# A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Unique Protocol ID:** SYNT001-103

NCT Number: NCT03075904

**Date of Protocol:** 18 September 2018

#### 1. PROTOCOL AND AMENDMENTS

- SYNT001-103 Protocol Version 1, 18 January 2017
- SYNT001-103 Protocol Amendment 1.1, 21 March 2017
- SYNT001-103 Protocol Amendment 1.1 SOC, 21 March 2017
- SYNT001-103 Protocol Amendment 2.0, 12 April 2017
- SYNT001-103 Protocol Amendment 2.0 SOC, 12 April 2017
- SYNT001-103 Administrative Letter 1.0, 10 May 2017
- SYNT001-103 Administrative Letter 2.0, 11 August 2017
- SYNT001-103 Administrative Letter 3.0, 21 September 2017
- SYNT001-103 Protocol Amendment 3.0, 10 October 2017
- SYNT001-103 Protocol Amendment 3.0 SOC, 10 October 2017
- SYNT001-103 Administrative Letter 4.0, 02 March 2018
- SYNT001-103 Protocol Amendment 4.0, 08 June 2018
- SYNT001-103 Protocol Amendment 4.0 SOC, 08 June 2018
- SYNT001-103 Protocol Amendment 5.0, 18 September 2018
- SYNT001-103 Protocol Amendment 5.0 SOC, 18 September 2018

### Syntimmune, Inc.

#### **CLINICAL STUDY PROTOCOL**

#### A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

**Medical Monitor:** PPD

**Original Protocol:** 

43 Thorndike Street, Cambridge, MA 01240

Phone: PPD extension PPD

Mobile: PPD

18 January 2017

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

**Confidentiality Statement** 

#### **SPONSOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the Investigator, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| PPD | |
|-----|--------------------------------|
| | 25/01/2017 |
| | Date of Signature (DD Mm YYYY) |

#### PROCEDURES IN CASE OF EMERGENCY

#### Serious Adverse Events

Any death, serious adverse event (SAE)\* occurring in a subject while receiving study drug or within 7 days of receiving study drug, even though the event may not appear to be study drug related, must be promptly reported (within 24 hours) by telephone or electronic communication to the sponsor (or designee).

#### **Emergency Contact Information**

| For SAE reporting: | | For any other q | | |
|---|---|---|---|---|
| Medpace Clinical Safety Medpace SAE hotline: Telephone: PPD PPD dial PP | dialP or PPD | PPD PPD Mobile phonePP Office phone: | D | ext.PPD |
| Facsimile: PPD | or PPD | | | |

#### **SAE CRITERIA**

- \* A <u>serious adverse event</u> (SAE) is any untoward medical occurrence that at any dose results in any of the following outcomes, regardless of relationship to study drug (see <u>Section 11.3.1</u>, Serious Adverse Events for additional information):
  - Death
  - Life-threatening adverse drug event
  - Inpatient hospitalization or prolongation of existing hospitalization
  - A persistent or significant disability/ incapacity
  - A congenital anomaly/birth defect
  - An important medical event that may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

Syntimmune, Inc.  Final 18 January 2017

#### **INVESTIGATOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the sponsor, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonization Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

Nothing in this document is intended to limit the authority of a physician to provide emergency

| edical care under applicable regulations. | |
|-------------------------------------------|--------------------------------|
| nvestigator Signature | Date of Signature (DD Mm YYYY) |
| ame of Investigator (please print) | |

#### 1 SYNOPSIS

| | A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus) |
|---|---|
| Protocol number | SYNT001-103 |
| Number of study centers | Approximately 10 (US) |
| Clinical phase | Phase 1b |
| | SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG immune complexes from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG containing immune complexes further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG immune complexes within and among compartments important in cellular immunity, it is further anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8+ and CD4+ T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG and IC that are involved in many autoimmune conditions and dismantle their ability to cause disease. SYNT001 targets mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP). While current treatments for certain autoimmune disorders including chronic steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are frequently associated with significant adverse effects, a |

| Study rationale | pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, leading to a significant decrease in total IgG, and thereby a corresponding decrease in the level of the pathogenic autoantibodies as well as the ICs to which they are associated, should lead to a decrease in the mucosal and cutaneous manifestations in subjects with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification. This study is being conducted to further evaluate the safety, tolerability, |
|---|---|
| | pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers. |
| Study objectives | Primary objective |
| | To evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus) |
| | Secondary objectives |
| | <ul> <li>To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels</li> <li>To assess the effect of 5 once-weekly doses of SYNT001 at different dose</li> </ul> |
| | levels on the following PD biomarkers: o Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM o Albumin |
| | To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers: |
| | o Serum anti-desmoglein (Dsg) (1 and 3) antibody levels |
| | o Pemphigus Disease Area Index (PDAI) |
| | To assess immunogenicity (anti-SYNT001 antibodies) |
| | Exploratory objectives |
| | To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including: |
| | <ul> <li>Serum anti-epithelial cell antibody (AECA) levels by indirect<br/>immunofluorescence</li> </ul> |
| | o Circulating immune complexes (CIC) |
| | o Complement component 3 (C3) |
| | <ul> <li>Exploratory biomarkers (FCGR2A (single nucleotide polymorphism-<br/>SNP), RNAseq, urine IgG)</li> </ul> |

# Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells

- o SYNT001 levels in skin biopsies (optional)
- To characterize corticosteroid use during the study

#### Study design

Phase 1b, multicenter, open-label, safety, tolerability, and activity study

#### Methodology

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of subjects | Dose |
|--------|-----------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs, and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All safety data and any available and relevant PD data through Day 42 (2 weeks after the last subject's last dose in Cohort 1) will be reviewed by a dose escalation committee before Cohort 2 is initiated. Escalation to Cohort 2 will proceed if there are no concerning safety signals and the review of available and relevant PD data supports advancing to a higher dose. The dose for Cohort 2 will be finalized after review of the safety and PD data, but will not exceed 30 mg/kg. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule as Cohort 1.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33 and 56. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, and 42 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects also will return to the clinic on Day 56 (28 days after receiving their last dose of study drug) for an End-of-Study/Follow-Up visit.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, adverse event (AE) assessments, concomitant medication assessments, and electrocardiograms (ECG).

#### **Number of subjects**

Approximately 16; two cohorts of 8 subjects each. An additional cohort of up to 8 subjects may be enrolled. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects with pemphigus foliaceus may be enrolled.

## Diagnosis and main entry criteria

#### **Inclusion criteria:**

Subjects must meet the following criteria to be included:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq$  18 years of age at the time of screening;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal:
  - c. History of at least one positive tissue-based test (e.g., biopsy, direct immunofluorescence [DIF])
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose
     12 months prior to screening;

- If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose
   (< 10% change in dose) for 6 weeks prior to screening;</li>
- c. If being treated with corticosteroids, must be  $\leq 1 \text{mg/kg/day}$  and stable (< 10% change in dose) for 2 weeks prior to screening;
- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 35.0 \text{ kg/m}^2$ ;
- 6. Has a negative urine pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through 60 days after the final study dose: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final study dose.

#### **Exclusion criteria:**

Subjects meeting any of the following criteria are to be excluded:

- 1. Subject unable or unwilling to comply with the protocol;
- Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG use within 60 days of screening;
- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;
- 8. Any exposure to an investigational drug or device within the 30 days prior to screening
- 9. Plasmapheresis or immunoadsorption within 60 days of screening

| | 10. Cellular therapy at any time prior to screening |
|---|---|
| | 11. Use of any immunosuppressive drugs apart from corticosteroids, |
| | azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of |
| | screening |
| | 12. Serum total IgG < 600 mg/dL; |
| | 13. Subject has any current medical condition that, in the opinion of the |
| | Investigator, may compromise their safety or compliance, preclude |
| | successful conduct of the study, or interfere with interpretation of the results |
| | (e.g., a significant pre-existing illness or other major comorbidity that the |
| | Investigator considers may confound the interpretation of the study results); |
| | 14. Any vaccination within 2 weeks of screening |
| Study drug, dosage, | SYNT001 |
| and administration | |
| | <b>Doses:</b> 10 mg/kg and 30 mg/kg. A third cohort of up to 8 subjects may be treated |
| | at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive. |
| | SYNT001 is provided as a liquid at a nominal concentration of 50 mg/mL. |
| | SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for |
| | infusion. |
| | Route of administration: IV in 250 mL over 1 hour |
| Control, dose, and | Not applicable |
| route of | |
| administration | |
| Duration of subject | Up to 70 days (10 weeks): Screening of up to 2 weeks (14 days); dosing period |
| participation and | of 4 weeks (28 days); and 4 weeks (28 days) of follow-up |
| duration of study | |

#### Prohibited Concomitant treatments

All treatments a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications may result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted.

Use of the following medications will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

#### Safety assessments

Safety assessments include AEs, serious adverse events (SAEs), PEs, vital sign measurements, clinical safety laboratory evaluations, ECGs, and reasons for treatment discontinuations due to toxicity. Safety assessments will be performed at specified time points and prior to discharge from the clinic. Vital sign measurements, including blood pressure, pulse rate, respiratory rate, and temperature will be monitored throughout the study. Pulse oximetry will be monitored during the study drug infusion and for 2 hours following the end of the infusion.

The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03) will be used for grading clinical and laboratory AEs.

| | The AE reporting period for a subject enrolled in the study begins when the subject provides informed consent and is continued for 28 days after the last dose of study drug. All AEs that occur in the enrolled subjects during the AE reporting period must be recorded, regardless of the relationship of the AE to study drug. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug should also be recorded. |
|---|---|
| Dose-escalation rules | Dose-limiting toxicity (DLT) will be defined generally as clinically significant, severe (Grade 3) AEs occurring in ≥ 2 subjects that are determined to be clinically significant and considered related to study drug. If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and no further dose-escalation will occur. If the dose-escalation stopping rule is met in Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics data will be reviewed and a cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met after Cohort 1 (10 mg/kg), dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met in Cohort 2, all safety data and all available pharmacodynamics data will be reviewed and a cohort may be added at a dose at least 30% lower than the Cohort 2 dose. If the stopping rule is not met after Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data. |
| Study stopping rule | If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, any further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the next appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects. |
| Individual stopping rule | Dosing for any individual subject will be discontinued (i.e., further treatment with the study drug will not be given) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator and Medical Monitor, suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject may be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a |

| | significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus. |
|---|---|
| Pharmacokinetics | The PK of SYNT001 will be evaluated following the first and last (fifth) doses of SYNT001. Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. Study drug concentration will be used to calculate the following PK parameters: $t_{1/2}$ , $C_{max}$ , $T_{max}$ , $AUC_{0-24}$ , and $AUC_{0-\infty}$ . |
| Pharmacodynamics/<br>Activity | PD samples will be collected for analysis of IgG (serial assessment of IgG levels to identify C <sub>min</sub> , T <sub>min</sub> ); IgG1-4 subtype levels; IgA levels; IgM levels; albumin levels; anti-Dsg (1 and 3) antibody levels; serum AECA by direct immunofluorescence; CIC; C3; exploratory biomarkers ( <i>FCGR2A</i> SNP, RNAseq, urine IgG, CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T, monocytes, NK cells and B cells). |
| Immunogenicity | Up to 4 samples will be collected for immunogenicity analyses. Samples will be collected on Days 0 (pre-dose), 14, 28, and 56. |
| Skin biopsy | Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33 and 56 to analyze SYNT001 levels. |
| Photography | Photographs of active lesions will be taken at Day 0. Follow-up photographs of the same areas will be taken on Days 33 and 56. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. |
| Statistical methods | Sample size consideration |
| | Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives. |
| | Data presentations/Descriptive statistics |
| | Three populations will be employed in the analysis of study data. |
| | The intent-to-treat (ITT) population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population. |
| | The PK population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters. |

• The PD population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the PK and ITT populations, where appropriate.

#### Criteria for evaluation

| Objective | Endpoint |
|---|---|
| Primary | |
| Safety and tolerability of 5 once- | AEs and clinical (safety) |
| weekly IV infusions of SYNT001 to | laboratory tests |
| subjects with pemphigus vulgaris or | |
| foliaceus | |
| Secondary | |
| PK of SYNT001 following a 1-hour IV | PK parameters: $t_{1/2}$ , $C_{max}$ , $T_{max}$ , |
| infusion | $AUC_{0-24}$ , and $AUC_{0-\infty}$ . |
| Effect of 5 once-weekly IV doses of | Changes in levels of IgG, IgG |
| SYNT001 on: | subtypes (IgG1-4), IgA, IgM, |
| • Total IgG (IgG1-4), IgA, IgM, and | albumin, serum anti-Dsg (1 and |
| albumin | 3) antibodies |
| • Serum anti-Dsg (1 and 3) antibodies | |
| Assess immunogenicity | Anti-SYNT001 antibodies |
| Disease Activity | PDAI Scores |
| Exploratory | |
| Effect of 5 once-weekly IV doses of | Changes in CIC; C3; AECA |
| SYNT001 on biomarkers including: | levels by indirect |
| • CIC | immunofluorescence; FCGR2A |
| • C3 | SNP; RNAseq; urine IgG, |
| <ul> <li>Serum anti-epithelial cell antibody</li> </ul> | CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T, |
| (AECA) levels | monocytes, NK cells and B |
| <ul> <li>Exploratory biomarkers (FCGR2A</li> </ul> | cells; urine IgG levels; changes |
| SNP, RNAseq, urine IgG) | in blood transcriptome |
| <ul> <li>Immune phenotyping by flow</li> </ul> | |
| cytometry | |
| Concomitant Treatment | Corticosteroid use during the |
| | study |
| SYNT001 levels in skin biopsies | Measures of SYNT001 levels in |
| • | skin biopsies |

Treatment-emergent AEs (TEAEs) will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred

term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, or treatment discontinuation will be listed by subject, and cohort using SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken, and outcome.

Laboratory results will be summarized by time point and cohort. The incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the central laboratory. Vital sign measurements will be summarized by cohort at each scheduled time point using descriptive statistics.

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and area under the curve (AUC). PK parameters will be determined using non-compartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

PD results will be summarized by cohort. Descriptive statistics of PD parameters for SYNT001 will include mean, SD, CV, median, minimum, and maximum.

Immunogenicity results will be summarized by cohort. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

**Table 1:** Study Assessments

| Timepoint (Study Day) | Screen<br>-14 to -1 | 0 | 1<br>(±1<br>hr) | 2<br>(± 2<br>hr) | 5 <sup>p</sup><br>(±4<br>hr) | 7<br>(±4<br>hr) | 12 <sup>p</sup><br>(±6<br>hr) | 14<br>(±6<br>hr) | 19 <sup>p</sup><br>(±6<br>hr) | 21<br>(±6<br>hr) | 28<br>(±6<br>hr) | 29<br>(±1<br>hr) | 30<br>(±2<br>hr) | 33<br>(±4<br>hr) | 42<br>(±3<br>day) | Follow-Up<br>56<br>(±5 days) or<br>ET Visit | Extended<br>Follow-<br>up <sup>q</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | | | | | | | | | | |
| Demographics/Medical History | X | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | | | | | | |
| Physical Examination <sup>a</sup> | X | X | | | | X | | X | | X | X | | | | X | X | |
| Vital Signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Pulse Oximetry <sup>c</sup> | | X | | | | X | | X | | X | X | | | | | | |
| Clinical Safety Labs <sup>d</sup> | X | X | | | | X | | X | | X | X | | | X | X | X | |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | | | | | | | | X | |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | |
| 12-Lead ECG <sup>f</sup> | X | X | | | | | X | | | | X | | | | | X | |
| Tetanus & VZV antibodies <sup>g</sup> | | X | | | | | | | | | | | | | | X | X |
| PDAI Score | | X | | | | X | | X | | X | X | | | X | X | X | |
| PK Sampling <sup>h</sup> | | X | X | X | X | | | | | | X | X | X | X | | | |
| Immunogenicity <sup>i</sup> | | X | | | | | | X | | | X | | | | | X | |
| Study Drug Administration <sup>j</sup> | | X | | | | X | | X | | X | X | | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4) <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| CIC | | X | | | X | X | X | X | X | X | X | | | X | X | X | |
| Anti-Dsg (1 & 3) antibody titer | X | X | | | | X | | X | | | X | | | X | | X | |
| C3 and AECA <sup>1</sup> | | X | | | | | | X | | | | | | X | | X | |
| FCGR2A <sup>m</sup> | | X | | | | | | | | | | | | | | | |
| RNAseq <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | |
| Urine IgG <sup>m</sup> | _ | X | | | | | | X | | | | | | X | | X | _ |
| Immune phenotyping <sup>n</sup> | | X | | | | | | | | | X | | | | | | |
| Optional Skin Biopsy | | X | X | X | | | | X | | | | | | X | | X | |
| Photography <sup>o</sup> | | X | | | | | | | | | | | | X | | X | |
| Adverse Events | | To be collected from the date that the ICF is signed until 28 days after last dose of study drug. | | | | | | | | | | | | | | | |
| Concomitant Medications | | To be collected from within 14 days prior to Day 0 through 28 days after last dose of study drug. | | | | | | | | | | | | | | | |

Concomitant Medications

To be collected from within 14 days prior to Day 0 through 28 days after last dose of study drug.

ECG = electrocardiogram; ET= Early Termination; HIV = human immunodeficiency virus; ICF = informed consent form; PD = pharmacodynamic; PK = pharmacokinetic; VZV = varicella-zoster virus

Syntimmune, Inc.  Final 18 January 2017

- a: Complete PE, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.
- b: **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. On Days 0, 7, 14, 21, and 28 vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- c: **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d: Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 6.7 for a complete list). Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42 and 56.
- e: **Pregnancy test:** To be performed at time of screening and prior to first dose of SYNT001 on Day 0 and on Day 56 (urine or serum test is acceptable, however, positive urine tests must be confirmed with serum testing.)
- f: Digital 12-lead ECG to be obtained after 5 minutes of rest in the supine position and in triplicate at least 1-2 minutes apart (see Section 6.6 for additional information). On Days 0 and 28 to be obtained 5 minutes after the completion of infusion. Day 12 ECG will be collected only if the visit is conducted at the study site.
- g: **Serology**: Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at 1 month after the Follow-Up visit (approximately 2 months after the subject's last dose); if still below the baseline value (or level of detection), the subject will be re-tested after another month (3 months after last dose). Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level on Day 56 and upon 2 retests (2 and 3 months following last dose of SYNT001), will be referred to their primary care physician for further management. See Section 6.7.3 for additional information.
- h: **PK:** Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. See Section 6.7.4 for additional information.
- i: Immunogenicity: Blood samples will be collected pre-dose when collected on dosing days. See Section 6.7.6 for additional information.
- j: Prior to **study drug infusion**, SYNT001 drug product is to be diluted in Dextrose 5% in Water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour using a 0.2-micron, inline filter. See Section 9 for additional information.
- k: Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, and IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 6.7.5 for additional information
- 1: Exploratory PD samples (C3 and AECA): collected pre-dose when collected on dosing days. See Section 6.7.5 for complete information.
- m: Samples to be collected and stored; pending review of clinical and pharmacodynamics assessments
- n: Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- o: Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 33 and 56. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- p: Visit Days 5, 12 and 19 may be conducted via at-home nursing in lieu of a subject visit to the study site.
- q: Extended follow-up visits will occur only if additional testing for anti-tetanus and/ or anti-VZV titers are required. These visits will occur as needed at approximately 2 months post last dose and 3 months post last dose.

Table 2: Timing Window Allowances for PK/PD Sampling, ECG, and Vital Sign Measurements

| Pharmacokinetic and Pharmacodynamic Sampling | |
|------------------------------------------------|--------------------|
| Timepoint | Tolerance Window |
| 0 hour | −240 min to 0 hour |
| 5 minutes post end-of-infusion | ± 5 minutes |
| 2, 4, & 6 hours post end-of-infusion | ± 15 minutes |
| 24 hours post end-of-infusion | ± 60 minutes |
| 48 hours post end-of-infusion | ± 120 minutes |
| ECG | |
| Timepoint | Tolerance Window |
| 5 minutes post end-of-infusion | ± 10 minutes |
| Vital Signs <sup>a</sup> | |
| Timepoint | Tolerance Window |
| 0 hour | −240 min to 0 hour |
| 15, 30, and 45 minutes after start of infusion | ± 5 minutes |
| 60 minutes after start of infusion | ± 10 minutes |
| 30, 60 and 120 minutes post end-of-infusion | ± 10 minutes |

a: Vital signs to include blood pressure, pulse rate, respiratory rate, oral temperature, and pulse oximetry.

#### TABLE OF CONTENTS

| PROCE | EDURES IN CASE OF EMERGENCY | 3 |
|--------|---------------------------------------------|----|
| INVEST | TIGATOR SIGNATURE | 4 |
| 1 SY | YNOPSIS | 5 |
| LIST O | F ABBREVIATIONS | 24 |
| 2 B | ACKGROUND AND RATIONALE | 26 |
| 2.1 | Study Rationale | 27 |
| 2.2 | Selection of Doses in this Study | |
| 2.3 | Compliance Statement | 28 |
| 3 S7 | TUDY OBJECTIVES | 29 |
| 3.1 | Primary Objective | 29 |
| 3.2 | Secondary Objectives | 29 |
| 3.3 | Exploratory Objectives | 29 |
| 4 S7 | TUDY DESIGN | 30 |
| 4.1 | Study Sites | 30 |
| 4.2 | Study Endpoints | 30 |
| 4.3 | Overview of Study Design | 31 |
| 4.4 | Randomization and Blinding | 33 |
| 5 S7 | TUDY POPULATION | 34 |
| 5.1 | Target Population | 34 |
| 5.2 | Inclusion Criteria | 34 |
| 5.3 | Exclusion Criteria | 35 |
| 6 S7 | TUDY PROCEDURES | 37 |
| 6.1 | Informed Consent | 37 |
| 6.2 | Demographics and Medical History | 37 |
| 6.3 | Physical Examination | 37 |
| 6.4 | Pemphigus Disease Area Index (PDAI) Scoring | 37 |
| 6.5 | Vital Sign Measurements | 37 |
| 6.6 | 12-Lead Electrocardiogram (ECG) | |
| 6.7 | Clinical Laboratory Measurements | |
| | 6.7.1 Pregnancy Testing | |
| | 6.7.2 Virology | 40 |

| | | 6.7.3 | Serum Tetanus Antibody and Varicella-Zoster Virus Antibody | • |
|---|---|---|---|---|
| | | 6.7.4 | Pharmacokinetics (PK) Sampling | |
| | | 6.7.5 | Pharmacodynamic Sampling | |
| | | 6.7.6 | Immunogenicity Testing | |
| | 6.8 | | y Drug Administration | |
| | 6.9 | | and Concomitant Medications | |
| | 6.10 | | erse Event Assessments | |
| | 6.11 | | ographs | |
| | 6.12 | Skin | Biopsy | 44 |
| 7 | ST | UDY A | SSESSMENTS | 45 |
| | 7.1 | Scree | ening Period: Day -14 to Day -1 | 45 |
| | 7.2 | Enro | Ilment and First Treatment: Day 0 | 45 |
| | 7.3 | Follo | ow-up: Day 1 | 47 |
| | 7.4 | Follo | ow-up: Day 2 | 47 |
| | 7.5 | Follo | ow-up: Day 5 | 48 |
| | 7.6 | Treat | ment Day 7 (Dose 2) | 48 |
| | 7.7 | Dose | 2 Follow-up Day 12 | 49 |
| | 7.8 | Treat | ment Day 14 (Dose 3) | 49 |
| | 7.9 | Dose | 3 Follow-up Day 19 | 51 |
| | 7.10 | Treat | ement Day 21 (Dose 4) | 51 |
| | 7.11 | Treat | ement Day 28 (Dose 5) | 52 |
| | 7.12 | Follo | ow-up Day 29 | 53 |
| | 7.13 | Follo | w-up Day 30 | 54 |
| | 7.14 | Follo | ow-up Day 33 | 54 |
| | 7.15 | Follo | ow-up Day 42 | 55 |
| | 7.16 | Follo | w-up Day 56 (End-of-Study) or Early Termination Visit | 55 |
| | 7.17 | Exte | nded Follow-up Visits | 56 |
| 8 | RE | MOVI | NG SUBJECTS FROM STUDY | 57 |
| | 8.1 | Subj | ect Withdrawal | 57 |
| | 8.2 | Stud | y Discontinuation | 58 |
| | 8.3 | Repl | acements | 58 |
| | 8.4 | Stop | oing Rule | 58 |
| | | 8.4.1 | Dose-Escalation Stopping Rule | 58 |
| | | 8.4.2 | Study Stopping Rule | 59 |
| | | 8.4.3 | Individual Stopping Rule | |
| 9 | ST | UDY D | RUG | 60 |
| | 9.1 | SYN | T001 | 60 |

Syntimmune, Inc.


Final 18 January 2017

| | 9.2 | Cohort | Dosing | 60 |
|---|---|---|---|---|
| | 9.3 | Timing | g of Dosing | 60 |
| | 9.4 | Identit | y of Investigational Products | 60 |
| | 9.5 | Investi | gational Product Retention at Study Site | 61 |
| | 9.6 | Warnii | ngs and Precautions | 61 |
| | | 9.6.1 | Infusion Reaction | 61 |
| | | 9.6.2 | Potential Immune Effects | 66 |
| 0 | CO | NCOMI | ΓANT MEDICATION AND TREATMENT | 67 |
| 1 | SA | FETY | | 69 |
| | 11.1 | Safety | Parameters | 69 |
| | 11.2 | Advers | se Event Definition | 69 |
| | 11.3 | Evalua | ting Adverse Events | 70 |
| | | 11.3.1 | Serious Adverse Events | 70 |
| | | 11.3.2 | Overdose | 71 |
| | | 11.3.3 | Non-Serious Adverse Events | 71 |
| | | 11.3.4 | Protocol-Related Adverse Events | 71 |
| | | 11.3.5 | Assessment of Causality | 71 |
| | | 11.3.6 | Recording Adverse Events | 72 |
| | | 11.3.7 | Planned Hospitalization | 72 |
| | | 11.3.8 | Reporting Pregnancies | 73 |
| | | 11.3.9 | Serious Adverse Event Reporting | 73 |
| | | 11.3.9.1 | Governing Regulatory Requirements | 73 |
| | | 11.3.9.2 | Time Frame for Reporting | 74 |
| | | 11.3.9.3 | Information to be Provided by the Investigator | 75 |
| | | 11.3.10 | Regulatory Reporting | 76 |
| | | 11.3.11 | Follow-up Information on a Serious Adverse Event (SAE) | 77 |
| | 11.4 | Other S | Safety Considerations | 77 |
| | | 11.4.1 | Laboratory Data | 77 |
| | | 11.4.2 | Medication Errors | 77 |
| | | 11.4.3 | Follow-Up of Adverse Events | 77 |
| | 11.5 | Safety | Monitoring for Dose Escalation | 78 |
| 12 | ST | ATISTIC | AL CONSIDERATIONS | 79 |
| | 12.1 | Genera | al Design | 79 |
| | 12.2 | | e Size Justification | |
| | 12.3 | - | cal Considerations | |
| | | 12.3.1 | Study Populations | 79 |
| | | 12.3.2 | Subject Accountability, Demographics, and Baseline Character | |

| | | 12.3.3 Concomitant Medications | 80 |
|----|------|-----------------------------------------------------|------|
| | 12.4 | Planned PK Analysis | 80 |
| | 12.5 | Safety Data | 81 |
| | 12.6 | Pharmacodynamic/Activity Data | 81 |
| | 12.7 | Immunogenicity Data | |
| | 12.8 | Interim Analysis | 82 |
| 13 | DA | TA QUALITY ASSURANCE | 83 |
| 14 | ST | UDY ADMINISTRATION | 84 |
| | 14.1 | Study Administrative Structure | 84 |
| | 14.2 | Ethical Conduct of the Study | 84 |
| | 14.3 | Informed Consent (ICF) | 84 |
| | 14.4 | Institutional Review Board | 85 |
| | 14.5 | Dose Escalation Committee | 85 |
| | 14.6 | Future Use of Subject Samples | 86 |
| 15 | CO | NDITIONS FOR MODIFYING THE PROTOCOL | 87 |
| 16 | CO | NDITIONS FOR TERMINATING THE STUDY | 88 |
| 17 | ST | UDY DOCUMENTATION, CRFS, AND RECORD KEEPING | 89 |
| | 17.1 | Investigator's Files and Retention of Documents | 89 |
| | 17.2 | Source Documents and Background Data | 89 |
| | 17.3 | Audits and Inspections | 90 |
| | 17.4 | Electronic Case Report Forms | 91 |
| 18 | MC | ONITORING THE STUDY | 92 |
| 19 | CO | NFIDENTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECORD | DS93 |
| 20 | PU | BLICATION OF DATA AND PROTECTION OF TRADE SECRETS | 94 |
| 21 | RF | FERENCES | 95 |

| T | IST | OI | $\mathbf{T}$ | ΛR | IFS |
|---|-----|----|--------------|----|-----|
| L | 451 | VΙ | 1 1 | ΑD | |

| Table 1: | Sable 1: Study Assessments | |
|---|---|---|
| Table 2: Timing Window Allowances for PK/PD Sampling, ECG, and Vi | | |
| | Measurements | 18 |
| Table 3: | Clinical Laboratory Panels | 39 |
| Table 4: | Pharmacodynamic/ Activity Assessments | 42 |
| Table 5: | Grading and Management of Allergic or Infusion-Related Reactions | 65 |
| Table 6: | Study Administrative Structure | |
| • | Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions. | |
| • | Anagement of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions Anagement of Severe (Grade 3 or higher) Infusion Reactions | |
| LICTOF | DRENDICEC | |
| | APPENDICES | |
| | A: NCI CTCAE, Version 4.03 | |
| Appendix E | 3: Pemphigus Disease Area Index | 97 |

#### LIST OF ABBREVIATIONS

ADA Anti-drug antibodies

AE Adverse event

AECA Anti-epithelial cell antibody
ALT Alanine aminotransferase
ANA Antinuclear antibody
AST Aspartate aminotransferase
ATC Anatomical therapeutic chemical

AUC<sub>0.24</sub> Area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose

 $AUC_{0-\infty}$  Area under the plasma concentration-time curve from pre-dose (time 0) to infinity

BLQ Below the limit of quantification

BMI Body mass index
BUN Blood urea nitrogen

CAR-T Chimeric antigen receptor and T-cell

CFR Code of Federal Regulations
C3 Complement component 3
CBC Complete blood count

CIC Circulating immune complexes

CIDP Chronic inflammatory demyelinating polyneuropathy

C<sub>max</sub> Maximum plasma concentration determined directly from the concentration-time profile

CRO Contract research organization

CV Coefficient of variation

CVID Common variable immune deficiency

DEC Dose escalation committee
D5W Dextrose 5% in Water
DIF Direct immunofluorescence
DNA Deoxyribonucleic acid
ECG Electrocardiogram

eCRF Electronic case report form
ESR Erythrocyte sedimentation rate
FcGR2a Fc Gamma R2a receptor
FcRn Neonatal Fc receptor

FDA Food and Drug Administration

GCP Good Clinical Practice

GI Gastrointestinal
HBV Hepatitis B virus
HCV Hepatitis C virus

HIPAA Health Insurance Portability and Accountability Act

HIV Human immunodeficiency virus

IB Investigator's brochure IC Immune complex

Pemphigus

ICF Informed consent form

ICH International Conference on Harmonization

IgA Immunoglobulin A
IgG Immunoglobulin G
IgG1-4 Immunoglobulin G1-G4
IgM Immunoglobulin M
IL-12 Interleukin 12

IND Investigational new drug
IRB Institutional review board

ITT Intent-to-treat
IUD Intrauterine devices

IV Intravenous

IVIG Intravenous immunoglobulin

MedDRA Medical Dictionary for Regulatory Activities

NHL Non-Hodgkin lymphoma
PD Pharmacodynamics
PE Physical examination
PK Pharmacokinetic
RBC Red blood cells
RNAseq RNA sequencing

QTcF Corrected QT interval using Fridericia's formula

SAE Serious adverse event
SAP Statistical analysis plan
SAS Statistical Analysis System

SD Standard deviation

SNP Single nucleotide polymorphism

SOC System Organ Class

SOP Standard operating procedures

SYNT001 A humanized, affinity matured IgG4-kappa monoclonal antibody

 $t_{1/2}$  Half-life

TEAE Treatment-emergent adverse event

T<sub>max</sub> Observed time to reach peak plasma concentration

TNF Tumor necrosis factor ULN Upper limit of normal

UNS Unscheduled

VZV Varicella-zoster virus

WAIHA Warm antibody autoimmune hemolytic anemia

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

#### 2 BACKGROUND AND RATIONALE

SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG ICs from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG-containing ICs further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen-presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG ICs within and among compartments important in cellular immunity, it is anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8<sup>+</sup> and CD4<sup>+</sup> T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG that are involved in certain autoimmune conditions and dismantle their ability to cause disease.

SYNT001 targets key mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP).

While current treatments for certain autoimmune disorders, including high-dose steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are associated with significant adverse effects, as well as delayed or non-durable responses.

Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies have been shown to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, which significantly decreases total IgG, including a corresponding decrease in the level of the pathogenic autoantibodies and the ICs to which they are associated, may lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification.

#### 2.1 Study Rationale

This study is being conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers.

#### 2.2 Selection of Doses in this Study

The planned dose levels of SYNT001 for this Phase 1b safety and proof-of-concept study of 10 mg/kg and 30 mg/kg were selected from careful review of the safety, tolerability, and PD effect on total IgG levels after single and repeat dosing of SYNT001 in non-human primates (NHPs), as well as the safety, tolerability, and PD effect on total IgG levels after single ascending doses of SYNT001 in healthy volunteers. In addition, further consideration was given to the desired level of FcRn blockade to achieve suppression of IgG to a range that has been previously correlated with disease remission. Further, we considered the potential effects of inhibiting FcRn function as they relate to immune complex associated innate and adaptive immunity in choosing these dose levels based upon exploratory studies of a single ascending dose of SYNT001 in healthy volunteers. From the NHP studies, single doses of SYNT001 produced a dose-dependent decrease in total IgG and a further decrease was seen with repeated weekly doses up to a maximum 70% reduction at 100 mg/kg. This magnitude of total IgG reduction is approaching the expected maximal effect of 100% inhibition of FcRn function based on murine studies also performed by Syntimmune and others [Roopenian 2003, Nixon 2015]. In the recently completed Phase 1a trial with SYNT001 in healthy volunteers a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the NHP studies further reductions are expected following multiple dosing. A comparable decrease in pathogenic autoantibodies is also anticipated.

In the NHP studies, relevant adverse effects, mild-to-moderate infusion reactions, were observed only after the third weekly IV administration, concurrent with the development of anti-SYNT001 antibodies. In the recently completed Phase 1a healthy male volunteer study, the doses of SYNT001 up to and including 30 mg/kg have been well tolerated. There were no dose limiting toxicities, serious adverse events, or any other safety concerns identified. No AEs were observed in the 1 and 3 mg/kg dose cohorts. A single Grade 2 AE was observed; a headache in the 10 mg/kg cohort, treated with acetaminophen. Other subjects had mild (Grade 1) AEs at 10 mg/kg. In Cohort 4 (30 mg/kg), 5 subjects received SYNT001. All five subjects experienced AEs; all were mild (Grade 1), transient and resolved spontaneously without intervention. Therefore, it is anticipated that the doses selected for this study should be well tolerated and have clinically relevant PD effects in patients with chronic pemphigus (vulgaris or foliaceus). For a summary of

findings from the single dose, clinical study in healthy subjects and further details on the nonclinical findings, please refer to the SYNT001 Investigator's Brochure.

#### 2.3 Compliance Statement

This study will be conducted in compliance with Good Clinical Practice (GCP), including the International Conference on Harmonisation (ICH) Guidelines and FDA regulations, consistent with the principles outlined in the Declaration of Helsinki. In addition, the Investigator agrees to adhere to all applicable local laws and regulatory requirements relevant to the use of new therapeutic agents.

The study will be conducted in compliance with the protocol. The appropriate Institutional Review Boards (IRBs) must approve the protocol, any amendments, and the subject informed consent form (ICF) prior to implementation.

Freely given written informed consent must be obtained from every subject prior to participation in this clinical trial. As part of this procedure, the Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or AEs that may occur. The study subject should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The Investigator or designee will provide the Sponsor with a copy of the IRB-approved informed consent form prior to the start of the study. The rights, safety, and well-being of participating subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (e.g., loss of medical licensure, debarment).

#### 3 STUDY OBJECTIVES

#### 3.1 Primary Objective

The primary objective of this study is to evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus).

#### 3.2 Secondary Objectives

The secondary objectives of this study are as follow:

- To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers:
  - o Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM
  - o Albumin
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers:
  - o Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
  - o Pemphigus Disease Area Index (PDAI)
- To assess immunogenicity (anti-SYNT001 antibodies)

#### 3.3 Exploratory Objectives

The exploratory objectives of this study are as follow:

- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including:
  - o Serum anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence
  - o Circulating immune complexes (CIC)
  - o Complement component 3 (C3)
  - Exploratory biomarkers (FCGR2A single nucleotide polymorphism-SNP, RNAseq, urine IgG)
  - Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
  - o SYNT001 levels in skin biopsies (optional)
- To characterize corticosteroid use during the study

#### 4 STUDY DESIGN

#### 4.1 Study Sites

This study will be conducted at approximately 10 sites in the United States (US).

#### 4.2 Study Endpoints

**Primary Outcome Measures:** Assessment of safety data (adverse events [AEs], serious adverse events [SAEs], vital sign measurements, ECGs and clinical laboratory tests) will be the primary safety measure.

#### **Secondary Outcome Measures**

#### Pharmacokinetics:

Half-life (t<sub>1/2</sub>), maximum plasma concentration determined directly from the concentration-time profile (C<sub>max</sub>), observed time to reach peak plasma concentration (T<sub>max</sub>), area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose (AUC<sub>0-24</sub>), and area under the plasma concentration-time curve from pre-dose (time 0) to infinity (AUC<sub>0-∞</sub>)

#### PD Biomarkers:

- Ig Assessments: Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o IgA levels
  - o IgM levels
- Albumin levels

#### Disease activity markers:

- Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
- Pemphigus Disease Area Index (PDAI) scores

#### Immunogenicity:

• Anti-SYNT001 antibodies

#### **Exploratory Outcome Measures**

Biomarkers, including:

- CIC
- C3
- Serum AECA levels
- Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG)

Syntimmune, Inc.  Final 18 January 2017

- Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- SYNT001 levels in skin biopsies (optional)

#### **Concomitant Treatments**

Corticosteroid use

Further details on the statistical and analytical plan for these endpoints are available in Section 12, Statistical Considerations.

#### 4.3 Overview of Study Design

This will be a multicenter, open-label study to assess the safety, tolerability, activity, PK, PD, and immunogenicity of 5 once-weekly IV infusions of SYNT001 to subjects with chronic pemphigus (vulgaris or foliaceus).

Planned doses of SYNT001 to be studied are 10 mg/kg and up to 30 mg/kg. Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 10 mg/kg or up to 30 mg/kg. Based on review of safety, PD, and clinical outcomes of the first cohort, the dose for the second cohort may be adjusted, but with a maximum dose of 30 mg/kg. Based on review of safety, PD and clinical outcomes from these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of<br>Subjects | Dose |
|--------|--------------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All data through Day 42

(2 weeks after the last subject's last dose in Cohort 1) will be reviewed before Cohort 2 is initiated. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule.

Safety evaluations will be conducted by a dose escalation committee (DEC). The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions. Dosing and dose escalation will proceed if the DEC has determined that it would be safe and appropriate to do so. In addition, over the course of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33 and 56. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, and 42 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects also will return to the clinic on Day 56 (28 days after receiving their last dose of study drug) for an End-of-Study/Follow-Up visit.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, AE assessments, concomitant medication assessments, and electrocardiograms (ECG).

Syntimmune, Inc.  Final 18 January 2017

**Note**: No vaccinations may be given from within 2 weeks of screening until 2 months following the last dose of study drug.

#### 4.4 Randomization and Blinding

This is an open-label study.

#### 5 STUDY POPULATION

#### 5.1 Target Population

This study will be conducted in approximately 16 male and female subjects (2 cohorts of 8 subjects each) with a confirmed diagnosis of pemphigus (vulgaris or foliaceus); however, a third cohort of up to 8 subjects may be added. Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through 28 days after their last dose. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects may be enrolled with pemphigus foliaceus.

#### 5.2 Inclusion Criteria

A subject must meet the following criteria to be eligible for the study:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq$  18 years of age;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal;
  - c. History of at least one positive tissue based test (biopsy, DIF)
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose > 12 months prior to screening;
  - b. If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
  - c. If being treated with corticosteroids, must be ≤ 1mg/kg/day and stable (< 10% change in dose) for 2 weeks prior to screening;
- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 35.0 \text{ kg/m}^2$ ;
- 6. Has a negative urine pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through 60 days after the final study dose: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final study dose.

### 5.3 Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

- 1. Unable or unwilling to comply with the protocol;
- Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG treatment within 60 days of screening;

- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;
- 8. Any exposure to an investigational drug or device within 30 days prior to screening;
- 9. Plasmapheresis or immunoadsorption within 60 days of screening
- 10. Cellular therapy at any time prior to screening
- 11. Use of any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of screening;
- 12. Serum total IgG < 600 mg/dL;
- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (e.g., a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results);
- 14. Any vaccination within 2 weeks of screening

#### 6 STUDY PROCEDURES

#### 6.1 Informed Consent

All subjects must take part in the informed consent process. Adequate time must be allowed for the subject to ask questions and make a voluntary decision. No protocol-specific procedures, including screening procedures, are to be performed until the subject has signed and dated an IRB-approved ICF. Subjects may withdraw consent at any time. Participation in the study may be terminated at any time without the subject's consent as determined by the Investigator.

### 6.2 Demographics and Medical History

Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and eCRF. Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery and concomitant treatments.

## 6.3 Physical Examination

A complete physical examination will be performed as outlined in Table 1. The complete PE will include measurements of weight (in kg) and height (in cm; height to be measured only at screening visit) and a review of the following body systems:

- General appearance
- Head, eyes, ears, nose, and throat
- Neck
- Respiratory
- Cardiovascular
- Abdomen
- Neurologic
- Extremities
- Dermatologic
- Lymphatic

Any abnormal and clinically significant findings from the PE must be recorded in the appropriate eCRF. Findings at screening and Day 0 (pre-dose) will be recorded as medical history.

### 6.4 Pemphigus Disease Area Index (PDAI) Scoring

Pemphigus severity and disease activity will be measured using the PDAI. See Appendix B.

#### 6.5 Vital Sign Measurements

Vital sign measurements will be collected after the subject has been sitting for 5 minutes. Vital sign assessments will include measurements of sitting blood pressure (mm Hg), heart rate (beats

per minute), respiration rate (breaths per minute), oral temperature (Celsius). Abnormal results are to be repeated after 5 minutes of rest. Pulse oximetry (%) also is to be measured. See Table 2 for timing window allowances with respect to measurement collection.

On Days 0, 7, 14, 21, and 28, vital sign measurements are to be obtained immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion. Details on the management of mild to moderate and severe infusion reactions can be found in Figure 1 and Figure 2. Abnormalities in vital sign measurements will be graded in severity per the NCI CTCAE scale Version 4.03.

Subjects should be seated quietly for at least 5 minutes in a chair with their backs supported, their feet flat on floor (legs uncrossed), and their arms bared on a hard surface, with the arm slightly abducted and bent, with palm up and the midpoint of upper arm at heart level. Correct cuff and bladder size should be utilized and the same cuff and arm should be used per subject throughout study.

## 6.6 12-Lead Electrocardiogram (ECG)

Digital 12-lead ECG measurements will be obtained at screening, on Days 0 and 28 at 5 minutes after the completion of the infusion and at the Day 56 (Follow-Up) Visit. Subjects who conduct their Day 12 visit at the investigative site, as opposed to an at-home nurse visit, will have an additional ECG performed. ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each 1 to 2 minutes apart. See Table 2 for timing window allowances with respect to performing ECG.

The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant.

Normal QTcF is  $\leq 450$  msec.

Abnormalities in the ECG that appear following therapy or that result in clinical signs and symptoms are considered clinically significant for the purposes of this study and will be recorded on the AE eCRF.

Syntimmune, Inc.  Final 18 January 2017

### 6.7 Clinical Laboratory Measurements

Collection time for all safety, PD, and exploratory labs are outlined in Table 1.

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and anti-drug antibody samples) will be performed using established methods by a central laboratory. Safety laboratory panels are defined as listed in Table 3. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and anti-drug antibody samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42 and 56. The total blood draw for each subject who completes the study at Day 56, will be approximately 308 mL. Please refer to the Laboratory Manual for more information.

**Table 3: Clinical Laboratory Panels** 

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| CBC with differential Erythrocyte Sedimentation Rate (ESR) | <ul> <li>Albumin</li> <li>Alkaline phosphatase</li> <li>ALT</li> <li>AST</li> <li>BUN</li> <li>Calcium</li> <li>Carbon dioxide</li> <li>Chloride</li> <li>Creatinine</li> <li>Glucose</li> <li>LDH</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total and direct bilirubin</li> <li>Total protein</li> <li>Uric acid</li> <li>C-Reactive Protein</li> </ul> | <ul> <li>Appearance</li> <li>Color</li> <li>pH</li> <li>Specific gravity</li> <li>Ketones</li> <li>Protein</li> <li>Glucose</li> <li>Nitrite</li> <li>Urobilinogen</li> <li>Blood/hemoglobin</li> <li>Leukocyte esterase</li> <li>Bilirubin</li> <li>Microscopic examination of sediment: only if the results of the urinalysis dipstick evaluation are positive for blood/hemoglobin</li> </ul> |
| Virology • Hepatitis C | | |
| Hepatitis B | | |

- HIV
- VZV
- Tetanus

ALT = alanine aminotransferase; AST = aspartate aminotransferase; CBC = complete blood count; BUN = blood urea nitrogen; HIV = human immunodeficiency virus; LDH = lactate dehydrogenase; VZV = varicella-zoster virus

Abnormalities in clinical laboratory tests that are considered clinically significant are to be recorded on the AE electronic case report form (eCRF) page. Laboratory results will be graded using the NCI CTCAE, Version 4.03. If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as an SAE (see Section 11.3.1).

#### 6.7.1 Pregnancy Testing

Pregnancy testing will be performed for women of childbearing potential at screening and prior to first dose of SYNT001 on Day 0 and Day 56 (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing.)

#### 6.7.2 Virology

Testing for HCV antibody, hepatitis B surface antigen, and HIV antibody will be performed at screening.

## 6.7.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

Samples for serum tetanus antibody and varicella-zoster virus antibody testing are to be collected at baseline (pre-dose, Day 0) and on Day 56 (Follow-Up visit). Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. Specifically, if the baseline VZV titer is above the detectable level, but tetanus is not, only the VZV antibody titer will be tested on Day 56. If the Day 56 results are below the baseline value, defined as greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at 1 month after the Follow-Up visit (approximately 2 months after the subject's last dose); if still below the baseline value (or level of detection), the subject will be re-tested after another month (3 months after last dose). Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level on Day 56 and upon 2 retests (2 and 3 months following last dose of SYNT001), will be referred to their primary care physician for further management.

### 6.7.4 Pharmacokinetics (PK) Sampling

Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. The actual time and date of each blood draw is to be recorded.

Study drug concentration will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-24}$ , and  $AUC_{0-\infty}$ .

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual

## 6.7.5 Pharmacodynamic Sampling

PD samples will be collected for analyses throughout the study. On Days 0, 7, 14, 21, and 28, samples should be collected prior to infusion of study drug. Measurements for albumin PD biomarkers will be derived from the clinical safety laboratory results. Samples for each type of PD will be collected according to the schedule shown in Table 4.

Table 4: Pharmacodynamic/ Activity Assessments

| Parameter | Collection Timepoints |
|---|---|
| IgG, IgG subtypes (IgG1-4), IgA, IgM | Screening, and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, and 56 |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, and 56 |
| • Albumin | Screening, and Days 0, 7, 14,21, 28, 33, 42, and 56 |
| Anti-Dsg (1 and 3) antibody titer | Screening, Days 0, 7, 14, 33, and 56 |
| <ul> <li>Complement component 3 (C3)</li> <li>Anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence</li> </ul> | Days 0, 14, 33, and 56 |
| Exploratory biomarker (RNAseq, Urine IgG) | Days 0, 14, 33, and 56 |
| Immune phenotyping by flow cytometry for<br>measurement of CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T,<br>monocytes, NK cells and B cells | Days 0 and 28 |
| Exploratory biomarker (FCGR2A SNP) | Day 0 |

See Table 2 for timing window allowances with respect to measurement collection. Detailed instructions for sample collection (including collection tubes) and preparation will be provided in a separate laboratory manual.

### 6.7.6 Immunogenicity Testing

Up to 4 serum samples will be collected for immunogenicity analyses. Samples will be collected on Days 0 (pre-dose), 14, 28, and 56.

SYNT001 is being developed for the acute and chronic therapy of autoimmune disorders. Although SYNT001 is a humanized IgG4 monoclonal antibody, exposure to SYNT001 in clinical trials could result in the development of anti-drug antibodies (ADAs), with potential consequences ranging from neutralization or lessening of drug efficacy to safety consequences such as allergic reactions. Testing will first detect binding ADAs, then, for all confirmed positive samples, there will be testing for neutralizing effects.

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

# 6.8 Study Drug Administration

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute IV infusions of SYNT001 10 mg/kg or up to 30 mg/kg. SYNT001 will be given as a 250-mL IV infusion over 1 hour using a 0.2-micron, inline filter. Based on review of safety data, as well as available and relevant PD results, and clinical outcomes of Cohort 1, a decision about proceeding with Cohort 2 will be made. Based on review of all safety data, available PD results, and clinical outcomes of these 2 cohorts, a third cohort of 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort No. | Study Drug | Dose Level<br>(mg/kg/dose) |
|------------|------------|----------------------------|
| 1 | SYNT001 | 10 mg/kg |
| 2 | SYNT001 | 30 mg/kg |

See Section 9.1 for dosing schedule.

#### 6.9 Prior and Concomitant Medications

All medications a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented on the source document and eCRF.

Note: No vaccinations may be given from within 2 weeks of screening until 2 months following the last dose of study drug.

#### 6.10 Adverse Event Assessments

Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form throughout their participation in the study, including a period of 28 days after study drug dosing. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE.

Clinical AEs will be graded using the NCI CTCAE, Version 4.03 (Appendix A).

**Note**: AEs resulting in a subject's permanent discontinuation from the study, regardless of seriousness or relationship to study drug, MUST be promptly reported to the sponsor. Additionally, subjects must be followed until return to normal and/or resolution of the AE.

Syntimmune, Inc.  Final 18 January 2017

See Section 11 for more information.

### 6.11 Photographs

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33 and 56. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

# 6.12 Skin Biopsy

Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33 and 56 to analyze SYNT001 levels.

#### 7 STUDY ASSESSMENTS

### 7.1 Screening Period: Day -14 to Day -1

Informed consent must be obtained before any study-specific samples are taken or study-specific tests or evaluations are conducted. The following assessments at the screening visit are to occur within 14 days before dosing. Study eligibility will be based on satisfying all the study inclusion and exclusion criteria.

At the screening visit, information will be collected and subjects will have clinical evaluations as follows:

- Informed consent (Section 6.1)
- Medical history and demographic data (Section 6.2)
- Review inclusion and exclusion criteria (Section 5.2, Section 5.3)
- Complete PE, including height and weight (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Section 6.6)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Hepatitis and HIV screen (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.2 Enrollment and First Treatment: Day 0

Study Day 0 is defined as the date the subject is administered their first dose of study drug. On Day 0, subjects will be asked to come to the clinic and the following procedures will be performed prior to the first dose of study drug:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)

- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody (Section 6.7)
- PDAI Score (Section 6.4)
- PK baseline sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - FCGR2A SNP
  - RNAseq
  - Urine IgG
  - Immune phenotyping
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral

Syntimmune, Inc.  Final 18 January 2017

temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)

- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.3 Follow-up: Day 1

On Day 1 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.4 Follow-up: Day 2

On Day 2 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.5 Follow-up: Day 5

On Day 5 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 0), subjects may return to the clinic or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.6 Treatment Day 7 (Dose 2)

On Day 7 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion

Syntimmune, Inc.  Final 18 January 2017

and at completion of the infusion (Section 6.5)

- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.7 Dose 2 Follow-up Day 12

On Day 12 ( $\pm$  6 hours) the subject may will return to the clinic, or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- If visit performed at the study site: 12-Lead ECG to be obtained in triplicate (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.8 Treatment Day 14 (Dose 3)

On Day 14 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)

Syntimmune, Inc.  Final 18 January 2017

- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.9 Dose 3 Follow-up Day 19

On Day 19 ( $\pm$  6 hours) the subject may return to the clinic, or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.10 Treatment Day 21 (Dose 4)

On Day 21,  $(\pm 6 \text{ hours})$  subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)

• AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.11 Treatment Day 28 (Dose 5)

On Day 28 ( $\pm$  1 Day), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (collected just prior to the start of the study drug infusion; record collection date and time for each PK sample) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Immune phenotyping
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion

Syntimmune, Inc.  Final 18 January 2017

- and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.12 Follow-up Day 29

On Day 29 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.13 Follow-up Day 30

On Day 30 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.14 Follow-up Day 33

On Day 33 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 28), subjects will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.15 Follow-up Day 42

On Day 42 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.16 Follow-up Day 56 (End-of-Study) or Early Termination Visit

On Day 56 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the sitting position) (Section 6.5)
- Serum tetanus antibody and VZV antibody; Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3

- AECA
- RNAseq
- Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.17 Extended Follow-up Visits

Extended follow-up visits will occur only if additional testing for anti-tetanus and/ or anti-VZV titers are required. These visits will occur as needed at approximately 2 months post last dose and 3 months post last dose. See Section 6.7.3.

#### 8 REMOVING SUBJECTS FROM STUDY

Every reasonable effort will be made to keep the subject in the study; however, if a subject is withdrawn from the study, every effort will be made by the Investigator to complete and report the reasons for withdrawal as thoroughly as possible. The reason(s) for termination must be clearly documented on the appropriate page of the eCRF. Once a subject discontinues from the study for any reason, every effort will be made to collect all clinical and laboratory data as scheduled for the Early Termination Visit (See Table 1). A termination eCRF must be completed for all enrolled subjects.

### 8.1 Subject Withdrawal

A subject's participation in the study may be prematurely discontinued for any of the following reasons:

- 1. The subject wishes to withdraw from the study.
- 2. Request by a regulatory agency (e.g., Institutional Review Board).
- 3. Subject experiences a significant or intolerable AE.
- 4. The subject experiences a significant adverse change in vital signs, PE findings, or a clinical laboratory parameter.
- 5. The subject has a need for a concomitant medication that is not permitted by the study protocol.
- 6. The subject experiences generalized impairment or mental incompetence that would result in the subject being unable to understand his or her participation in the study.
- 7. If, in the Investigator's medical judgment, further participation would be injurious to the health and well-being of the subject, or is not in the best interest of the subject.
- 8. Administrative reasons, such as subject non-compliance or a major protocol violation.

Subjects who are withdrawn from this study due to an AE determined to be related to study drug are to be followed until there is either:

- Resolution or stabilization of the AE determined to be related
- The subject is lost to follow-up
- The event is otherwise explained

If there is a persistent AE contributing to discontinuation that is determined to be related to SYNT001, subjects must be followed with appropriate medical management until resolution or stabilization.

A reasonable effort should be made to contact any subject lost to follow-up during the study to complete assessments and retrieve any outstanding data. If the subjects are unreachable by telephone after three (3) attempts, the minimum of a registered letter should be sent requesting that contact be made with the Investigator to report survival information.

#### 8.2 Study Discontinuation

Syntimmune Inc. has the right to terminate or to stop the study at any time. Reasons for study discontinuation may include, but are not limited to the following:

- The incidence or severity of AEs in this or other related studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Drug supply issues
- Excessive subject self-withdrawal
- Significant protocol violations (e.g., violation of eligibility criteria, dosing errors, missing data for study endpoint analysis)

### 8.3 Replacements

Enrolled subjects withdrawn for a reason other than an AE will be replaced if they have not been dosed or have only received one dose of study drug at the time of discontinuation, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through 28 days after their last dose.

#### 8.4 Stopping Rule

# 8.4.1 Dose-Escalation Stopping Rule

Dose-limiting toxicity (DLT) will be defined generally as clinically significant, severe (Grade 3) AEs occurring in  $\geq$ 2 subjects that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and no further dose-escalation will occur. If the dose-escalation

Syntimmune, Inc.  Final 18 January 2017

stopping rule is met in Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics will be reviewed and a cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met after Cohort 1, dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met in Cohort 2, all safety data and all available pharmacodynamics will be reviewed and a cohort may be added at a dose a minimum of 30% lower than the Cohort 2 dose. If the stopping rule is not met after Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data.

#### 8.4.2 Study Stopping Rule

If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects.

# 8.4.3 Individual Stopping Rule

Dosing for any individual subject will be discontinued (i.e., no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator and Medical Monitor suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject may be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus.

#### 9 STUDY DRUG

For detailed information regarding SYNT001 preparation and administration, refer to the Pharmacy Manual.

#### 9.1 SYNT001

SYNT001 is provided in vials containing 5 mL SYNT001 (extractable volume) at a nominal concentration of 50 mg/mL. The product is supplied as a liquid at pH  $6.5 \pm 0.5$ . SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for infusion. SYNT001 will be infused via IV in 250 mL over 1 hour using a 0.2-micron, inline filter.

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these two cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

The specification for host cell DNA in SYNT001 is < 2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing is limited to 5000 mg of SYNT001. Therefore, at the highest dose possible in this study (45 mg/kg), maximum subject weight will be limited to 111 kg.

### 9.2 Cohort Dosing

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. Cohort 2, and Cohort 3 if added, will be dosed per the same schedule

#### 9.3 Timing of Dosing

On Days 0, 7, 14, 21, and 28, subjects will receive a 60-minute IV infusion of SYNT001 in the morning. The date and time the dose is administered will be recorded.

#### 9.4 Identity of Investigational Products

All supplies of SYNT001 will be supplied by Syntimmune and must be stored refrigerated (2°C to 8°C/36°F to 46°F) in the carton and protected from light, in a securely locked area, accessible to authorized persons only, until needed for dose preparation. Qualified site personnel will

Syntimmune, Inc.  Final 18 January 2017

inventory the investigational product received and will maintain records of disposition of the drug, including dates, quantity and use.

# 9.5 Investigational Product Retention at Study Site

The Investigator (or designee) is responsible for maintaining accurate accountability records of the investigational product throughout the clinical study. All study drug received at the site must be inventoried and accounted for in an accountability log provided by the Sponsor. All dispensing and accountability records will be available for Sponsor review. Study drug accountability will be verified during on-site monitoring visits.

Upon the completion or termination of the study, and upon written authorization from the Sponsor, or its representative, all unused and/or partially used study drug should be returned or destroyed at the investigational site, as specified by Sponsor. It is the Investigator's responsibility to ensure that the Sponsor, or its representative, has provided written authorization that procedures for proper disposal of the study drug have been established, and that appropriate records of the disposal are documented and maintained. No unused study drug may be disposed until fully accounted for by the Sponsor monitor (or designee)

## 9.6 Warnings and Precautions

**Note:** Subjects must not receive any vaccinations from within 2 weeks of screening until 2 months after the last dose of study drug.

#### 9.6.1 Infusion Reaction

SYNT001 will be given as an IV infusion over 1 hour. As with all mAbs administered by IV infusion, infusion reactions are possible. In nonclinical testing of SYNT001 in NHPs, clinical observations were limited to infusion reactions due to the immunogenicity of SYNT001 in NHPs. These reactions included transient emesis/vomitus which typically occurred within 1 hour of dosing at all dose groups, but only after the third weekly infusion following the development of ADAs. Transient histamine-type responses were noted 30 minutes post-dose in some animals in all dose groups, but only following the third weekly infusion as above. These reactions were consistent with a histamine reaction (decreased activity, periocular swelling, erythema, facial flushing, eyelids partially/completely closed, and/or generalized weakness). With the exception of vomitus/emesis and red skin discoloration associated with injection or blood draw sites, these observations spontaneously resolved within 1-hour post-dose. Subsequent pretreatment with intramuscular diphenhydramine prevented further histamine-type reactions. All doses of SYNT001 were administered by bolus infusion over approximately 5 minutes in the NHP

studies. However, all of the observed infusion reactions (including vomitus/emesis and histamine-type reactions) associated with ADAs are not at all predictive of what may occur in humans [Bugelski 2004, Ponce 2009] and furthermore, are not considered relevant to predicting responses in humans [ICH S6(R1) 2011].

Typically, infusion reactions to monoclonal antibodies observed in human studies develop within 30 minutes to 2 hours after the initiation of drug infusion, although symptoms may be delayed for up to 24 hours. Most are mild in severity, although severe and even fatal reactions can occur.

## Guidelines for Grading and Management of Allergic or Infusion-Related Reactions

Allergic and/or infusion-related reactions include hypersensitivity reactions and cytokine release syndromes. These reactions are experienced by patients during or within hours of the infusion of monoclonal antibody therapy. Symptoms can include flushing, alterations in heart rate and blood pressure, dyspnea, bronchospasm, back pain, fever, urticaria, edema, nausea, and all types of rashes. Anaphylaxis is recognized as a severe, life-threatening, generalized, or systemic reaction. This is a medical emergency characterized by rapidly developing life-threatening airway and/or breathing and/or circulation problems usually associated with skin or mucosal changes.

Management of Grade 1 infusion reactions include decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen.

Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. See Figure 1 and Figure 2 for details on the management of Grades 1-2 and Grade 3 or higher infusion reactions. The severity of and management of allergic or infusion-related reactions will be graded and managed using NCI CTCAE Version 4.03 (see Table 5).

Figure 1: Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions



If symptoms and signs resolve completely either spontaneously or after administration of diphenhydramine with or without hydrocortisone, consider rechallenge:

Wait at least 20 minutes following medication administration before commencing rechallenge at an infusion rate of 50% or less of the initial infusion rate or

Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction

Syntimmune, Inc.  Final 18 January 2017

Figure 2: Management of Severe (Grade 3 or higher) Infusion Reactions

Subject presents with any of the below:

- Urticaria
- Airway threatened by angioedema
- Angioedema: Lip, mouth, facial swelling
- Respiratory compromise wheezing, dyspnea, stridor or hypoxia (O2 saturation < 90%)
- BP < 90 mmHg SBP or >30% decrease from patient baseline



Start basic life support:

- High oxygen flow
- On bed, head down, legs up
- Large bore IV cannula, 1 L normal saline STAT
- Initiate vital signs at least every 15 minutes



Consider (under medial direction):

Epinephrine 1:1000

• 0.3 mg (0.3 mL) IM into lateral thigh



Airway Threatened: Nebulized epinephrine 1:1000, 3–5 mL (3–5 mg)

**Bronchospasm:** Nebulized salbutamol 5 mg

(Wheeze or Hypoxia) Consider: Intubation / nebulized epinephrine

**Hypotension:** Place on cardiac monitor

(Systolic BP <100 mmHg) Further epinephrine 1:1000, 0.3 mg IM and

IV normal saline bolus 20 mL/kg STAT as needed

Have vasopressin on hand



Transfer to Emergency Room/ICU Observe until all symptoms resolved.

Table 5: Grading and Management of Allergic or Infusion-Related Reactions

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Infusion-<br>Related<br>Reaction | Mild transient<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Allergic<br>Reaction | Transient<br>flushing or<br>rash, drug<br>fever<br>< 38.0°C.<br>Intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Anaphylaxis | - | - | Symptomatic<br>bronchospasm, with or<br>without urticarial;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Cytokine<br>release<br>syndrome | Mild<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>pressor or<br>ventilator<br>support<br>indicated | Death |

Abstracted from NCI CTCAE Version 4.03.

### 9.6.2 Potential Immune Effects

An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels after a single dose and further decreases after multiple doses up to a 70% to 80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within normal limits occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.

Given the normal adult range of IgG of 700 to 1600 mg/dL (in some references), with a mean of 1150 mg/dL, a 50% decrease in the mean would be to 575 mg/dL and a 50% decrease from the low end of the normal range of 700 mg/dL would be to 350 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 140 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency [Ameratunga 2013], the levels will be transient. Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to reverse the low IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

An antibody blocking FcRn is expected to also down modulate innate and adaptive immunity and the catabolism of IgG-containing immune complexes (IC). Specifically, it is expected that anti-FcRn will promote the clearance of IgG-containing ICs and the effects of these IC on stimulating innate immune cell production of inflammatory cytokines (e.g., IL-12, interferon-γ, and tumor necrosis factor [TNF]) and inhibit the processing and presentation of antigens contained within IC and thus the antigen-specific activation of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells. Therefore, subjects with pre-existing conditions that are dependent upon IgG antibodies, such as chronic infections (e.g., HIV, HBV or HCV), will be excluded from this study, as will subjects with active infection in general.

SYNT001 administration could decrease the level of protective antibodies from prior vaccinations. Protective antibody levels for tetanus and varicella-zoster virus (chickenpox) are to be tested in accordance with Section 6.7.3.

#### 10 CONCOMITANT MEDICATION AND TREATMENT

All treatments a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications may result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted

Use of the following treatments will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine.
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

In cases in which concomitant medications are used, details to be recorded include the following: medication name, start date and time, stop date and time, dose, route, frequency, and reason for use. The concomitant medication names are to be coded using the World Health Organization

(WHO) Drug Dictionary (WHO-DD March 2013, Type B2 or later) and classified by anatomical therapeutic chemical (ATC) categories.

 Final 18 January 2017 Syntimmune, Inc. 

#### 11 SAFETY

### 11.1 Safety Parameters

Clinical and laboratory AEs will be graded using the NCI CTCAE; Version 4.03 (See Appendix A).

Subjects will be monitored throughout the treatment and follow-up period for occurrence of AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status, vital sign measurements, and laboratory data (including PD). Safety parameters to be measured/assessed include PEs, vital sign measurements, hematology, serum chemistries, urinalysis, and ECG.

#### 11.2 Adverse Event Definition

An AE is defined as any untoward medical occurrence in a clinical trial subject associated with the use of a drug, whether considered drug related. An AE can be an unfavorable and unintended sign (e.g., an abnormal laboratory value finding), a symptom, or a disease temporally associated with the use of a drug, without judgment as to causality. An AE can arise from use of the drug (e.g., use in combination with another drug) and from any route of administration, formulation or dose, including an overdose. An AE also includes, but is not limited to, any clinically significant worsening of a pre-existing condition. Examples include:

- Any sign, symptom, physical finding, or laboratory result that has worsened in nature, severity or frequency compared to baseline;
- Reactions from an investigational drug, including those occurring because of an overdose, abuse of the study drug, withdrawal phenomena, sensitivity or toxicity;
- Concurrent illness that was not present or worsens in nature, severity, or frequency compared to baseline;
- Injury or accident; and/or
- Exacerbation of a pre-existing condition.

For data collection, all untoward events that occur after informed consent through 28 days after study drug dosing are to be recorded on eCRFs by the investigational site.

While pregnancy alone is not considered as an AE or SAE, any pregnancy complication(s) should be recorded as an AE(s) or SAE(s) (if applicable). Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions (see below). Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. If a female subject becomes pregnant during the conduct of the study, the Investigator must notify the Sponsor according to the procedures provided in Section 11.3.8).

## 11.3 Evaluating Adverse Events

The Investigator will determine the seriousness, intensity, and causality of an AE associated with the use of the study drug (i.e., events where there is a reasonable possibility that the event may have been caused by the study drug) based on the definitions that follow.

#### 11.3.1 Serious Adverse Events

(Notify Medpace Safety within 24 hours; document on eCRF)

The SAE definition and reporting requirements are in accordance with Title 21 Part Code of Federal Regulations (CFR) 312.32 and the Guidance for Industry and Investigators Safety Reporting Requirements for Investigational New Drug (INDs) and Bioavailability /Bioequivalence Studies.

SAE: An AE is considered "serious" if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:

• <u>Death:</u> This includes any death that occurs while the subject is "on study" as well as any death that occurs within 28 days after study drug administration.

**Note:** Death is an outcome of an AE, and not an AE. The event(s) that caused death (e.g., illness, accident) is the SAE. Death due to any other cause(s) must also be reported as an outcome of the reportable SAE.

- <u>Life-threatening adverse drug event:</u> An AE or suspected adverse reaction is considered "life threatening" if, in the view of either the Investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.
- Inpatient hospitalization or prolongation of existing hospitalization:

In the absence of an AE, the Investigator should not report hospitalization or prolongation of hospitalization. This is the case in the following situations:

- Hospitalization or prolongation of hospitalization is needed for a procedure required by the protocol
- Hospitalization or prolongation of hospitalization is part of routine procedure followed by study center
- Hospitalization for survey visits or annual physicals
- Hospitalization for observation with release within 24 hours

In addition, a hospitalization planned before the start of the study for a pre-existing condition, which has not worsened, does not count as an SAE.

# • Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

- Congenital anomaly/birth defect
- <u>Important medical event:</u> An event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 11.3.2 Overdose

An overdose is defined as a significant variation from the recommended/scheduled dosage for a product. The dosing for this study will be conducted in a controlled clinical setting and an overdose is not anticipated. However, in the event of an accident, for this study, an overdose of SYNT001 is considered a dose that is two-fold higher than the intended dose for the subject.

#### 11.3.3 Non-Serious Adverse Events

(Document on eCRF)

All other AEs, not fulfilling the previous definitions, are classified as non-serious.

#### 11.3.4 Protocol-Related Adverse Events

AEs that are not test drug related may nevertheless be considered by the Investigator or the Medical Monitor to be related to the conduct of the clinical study. That is, the event may be related to the fact that a subject is participating in the study. For example, a protocol-related AE may be an event that occurs during a screening period or that is related to a procedure required by the protocol.

#### 11.3.5 Assessment of Causality

A medically qualified Investigator must assess the relationship of any AE (including SAEs) to the use of the investigational product, as related or not related, based on clinical judgment and using all available information, and may include consideration of the following factors:

- Possible alternative causes of the AE, including the disease under treatment, pre-existing conditions, concomitant use of other drugs, and presence of environmental or genetic factors.
- The temporal association between drug exposure and onset of the AE.
- Whether the manifestations of the AE are consistent with known actions or toxicity of the investigational product.
- The AE resolved or improved with decreasing the dose or stopping use of the investigational product (dechallenge). Judgment should be used if multiple products are discontinued at the same time.

The causal relationship between the study medication and the AE will be assessed using one of the following categories:

**Not Related:** Factors consistent with an assessment of Not Related include:

- Temporal relationship is lacking (e.g., the event did not occur within a reasonable time frame following administration of the study medication); or
- Other causative factors more likely explain the event (e.g., a pre-existing condition, other concomitant treatments).

**Related:** Factors consistent with an assessment of Related include:

• There is a positive temporal relationship (e.g., the event occurred within a reasonable time frame following administration of study medication); or

The AE is more likely explained by the investigational product than by another cause (i.e., the AE shows a pattern consistent with previous knowledge of the investigational product or the class of the investigational product)

#### 11.3.6 Recording Adverse Events

All AEs (including SAEs) are to be accurately recorded on the <u>Adverse Event</u> page of the subject's eCRF. The severity of each AE will be graded using the NCI CTCAE, Version 4.03. The date of onset as well as the end date of the event also should be recorded or the event should be entered as "ongoing". In addition, the method used to treat the AE and the outcome of the AE also will be noted. The Investigator will assess the relationship of the event to study drug.

#### 11.3.7 Planned Hospitalization

A hospitalization planned by the subject prior to the first dose of study medication is considered a therapeutic intervention and not the result of a new SAE and should be recorded as medical

Syntimmune, Inc.  Final 18 January 2017

history. If the planned hospitalization or procedure is executed as planned, the record in the subject's medical history is considered complete. However, if the event/condition worsens during the trial, it must be reported as an AE.

#### 11.3.8 Reporting Pregnancies

If a female subject or the female partner of a male subject becomes pregnant during the course of the study, the Investigator must report the pregnancy to the Medpace Safety using the **Pregnancy Reporting Form** within **24 hours** of becoming aware of the event. The Investigator must obtain consent to collect pregnancy information (including the status of the newborn, if applicable).

If some of the information required for completion of the Pregnancy Reporting Form is unavailable at the time of the initial report, follow-up reports will be completed and submitted within 24 hours of becoming aware of the new information. Any pregnancy will be followed through delivery for the observation of any SAEs. Any SAE that occurs during pregnancy must be recorded on the SAE report form in the EDC system (e.g., maternal serious complications, therapeutic or spontaneous abortion, ectopic pregnancy, stillbirth, neonatal death, congenital abnormality, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs (See Section 11.3.9).

#### 11.3.9 Serious Adverse Event Reporting

#### 11.3.9.1 Governing Regulatory Requirements

Compliance with this request for prompt reporting is essential in that the sponsor is responsible for informing the US Food and Drug Administration (FDA) and other regulatory authorities as well as all other participating Investigators of the event.

Under FDA ruling (US Code of Federal Regulations, Title 21 CFR Part 312.32) and the ICH Guidelines for Clinical Safety Data Management Definitions and Standards for Expedited Reporting, the sponsor is required to submit written documentation, in the form of a safety report, detailing:

- Any event associated with the use of the drug, that is both serious and unexpected, or
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects, including reports of <u>mutagenicity</u>, <u>teratogenicity</u>, <u>or carcinogenicity</u>.

Written submission must be made by the sponsor to the FDA and the IRBs as soon as possible and in no event later than 15 calendar days after the sponsor's initial notification of the event. The sponsor shall also inform all Investigators.

#### 11.3.9.2 Time Frame for Reporting

Any death, SAE, pregnancy, or unexpected (and severe) AE experienced by the subject after informed consent or within 28 days of receiving study drug, regardless of relationship to study drug, or any death that occurs more than 28 days after receiving study drug, and is believed to be study drug related, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee).

Contact information for **SAE** reporting:



Additionally, the Investigator will be able to contact the **Medical Monitor**:



#### 11.3.9.3 Information to be Provided by the Investigator

SAEs must be recorded on the SAE form in the EDC system. This requirement includes all SAEs that occur after informed consent and through 28 days after study drug dosing, and in addition, any SAE that are assessed as related to study treatment by the Investigator, even if the SAE occurs more than 28 days after study drug dosing.

The minimum information required for SAE reporting includes identity of Investigator, site number, subject number, an event description, SAE term(s), onset date, the reason why the event is serious (i.e., the seriousness criteria) and the Investigator's assessment of the relationship of the event to study treatment. Additional SAE information including medications or other therapeutic measures used to treat the event, action taken with the study treatment due to the event, and the outcome/resolution of the event will be recorded. Paper forms for reporting SAEs will be provided to the study sites as back-up in case the EDC system is not accessible.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. Furthermore, the Investigator may be required to provide supplementary information as requested by Syntimmune or designee.

Syntimmune, Inc.  Final 18 January 2017

When reporting an SAE, the following additional points should be noted:

- When the diagnosis of an SAE is known or suspected, the Investigator should report the
  diagnosis or syndrome as the primary SAE term, rather than as signs or symptoms. Signs
  and symptoms may then be described in the event description. For example, dyspnea
  should not be used as an SAE term if the diagnosis, which caused the dyspnea, is known
  to be malignant pleural effusion.
- Death should not be reported as an SAE, but as an outcome of a specific SAE, unless the event preceding the death is unknown. In the exceptional case where the events leading to death are unknown, then death may be used as an event term. If an autopsy was performed, the autopsy report should be provided.
- While most hospitalizations necessitate reporting of an SAE, some hospitalizations do not require SAE reporting, as follows:
  - Elective or previously scheduled surgery, e.g., a previously scheduled ventral hernia repair
  - Procedures for pre-existing conditions that have not worsened after initiation of treatment
  - Pre-specified study hospitalizations for observation
  - Events that result in hospital stays of less than 24 hours and that do not require admission, e.g., an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics
- SAEs must, however, be reported for any surgical or procedural complication resulting in prolongation of the hospitalization.

#### 11.3.10 Regulatory Reporting

Syntimmune (or designee) will process and evaluate all SAEs as soon as the reports are received. For each SAE received, Syntimmune will decide as to whether the criteria for expedited reporting have been met.

Syntimmune (or designee) will submit SAEs that meet the criteria for expedited reporting to the regulatory authorities in accordance with local regulations governing safety reporting. Reporting of SAEs by the Investigator to his or her IRB will be done in accordance with the standard operating procedures and policies of the IRB. Adequate documentation must be maintained showing that the IRB was properly notified.

#### 11.3.11 Follow-up Information on a Serious Adverse Event (SAE)

Appropriate diagnostic tests should be performed and therapeutic measures, if indicated, should be instituted. Appropriate consultation and follow-up evaluations should be carried out until the event has returned to baseline or is otherwise explained by the Investigator.

If all required information on the SAE form is not available at the time of the initial report, follow-up information will be completed in the EDC system.

#### 11.4 Other Safety Considerations

#### 11.4.1 Laboratory Data

All laboratory data obtained during the study should be reviewed. Any abnormal value that leads to a change in subject management (e.g., requirement for additional medication or monitoring) or is of clinical significance by the Investigator should be reported as an AE and/or SAE as appropriate, unless this value is consistent with values obtained before entry into the study.

#### 11.4.2 Medication Errors

Any medication error that results in an AE, even if it does not meet the definition of serious, requires reporting within 24 hours to the safety Medical Monitor.

#### 11.4.3 Follow-Up of Adverse Events

Any SAE or AE assessed as related that led to treatment discontinuation (including clinically significant abnormal laboratory values that meet these criteria) and ongoing 28 days after study drug dosing must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. This follow-up guidance also applies to related SAE that occur more than 28 days after study drug dosing. The status of all other continuing AEs will be documented as of 28 days after study drug dosing. The Investigator will follow all subjects who experience AEs until there is a return to the subject's baseline condition, or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary.

Where a diagnosis is possible, it is preferable to report this diagnosis rather than a series of terms (signs/symptoms) relating to the diagnosis.

#### 11.5 Safety Monitoring for Dose Escalation

Following dosing in each cohort, all safety/tolerability data (e.g., PEs, vital signs [including pulse oximetry], clinical safety laboratory tests, ECGs and AE/SAE assessments) as well as any available and relevant PD data collected through Day 42 will be reviewed by the DEC. A decision to escalate to the next cohort will be made. The recommendation may be to continue to the next scheduled dose level, discontinue the study or to modify dosing to a dose less than the current dose or higher than the current dose but lower than the next planned dose.

#### 12 STATISTICAL CONSIDERATIONS

All descriptive and inferential statistical analyses will be performed using the most recently released and available Statistical Analysis System (SAS) software, unless otherwise noted. Missing data will not be imputed unless otherwise stated. All clinical data captured will be provided in data listings. A Statistical Analysis Plan (SAP) and a Pharmacokinetic Analysis Plan (PAP) will be finalized prior to database lock.

#### 12.1 General Design

All data for enrolled subjects will be presented in data listings by subject number.

Continuous data will be described using descriptive statistics: number of observations (n), mean, standard deviation (SD), median, minimum, and maximum. Frequencies and percentages will be used for summarizing discrete (categorical) data. When categorical data are presented, the percent will be suppressed when the count is zero to draw attention to the non-zero counts. The denominator for all percentages, unless otherwise specified, will be the number of subjects in the specified analysis population.

#### 12.2 Sample Size Justification

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

#### 12.3 Statistical Considerations

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). The SAP may modify the plans outlined in the protocol; any deviations from the previously described statistical plan will be described and justified in an SAP amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate and will be described in the SAP. Methods of handling of missing data for different endpoints will be further specified in the SAP. In general, where individual data points are missing because of insufficient samples, dropouts, or other reasons, the data will be analyzed based on reduced denominators unless specified otherwise in the SAP.

Results will be summarized by cohorts.

### 12.3.1 Study Populations

Three populations will be employed in the analysis of study data:

Syntimmune, Inc.  Final 18 January 2017

- The **intent-to-treat (ITT)** population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population.
- The **PK** population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters.
- The **PD** population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the ITT, PK, and PD populations, where appropriate.

#### 12.3.2 Subject Accountability, Demographics, and Baseline Characteristics

Subject disposition, demographic information and baseline characteristics will be presented. Any discrepancy between treatment to be given and treatment received will be accounted for in these displays.

#### 12.3.3 Concomitant Medications

Concomitant medications will be coded using WHO Drug Dictionary (WHO-DD March 2013, Type B2 or later) and the data will be summarized and presented in tables and listings.

#### 12.4 Planned PK Analysis

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and  $AUC_{0-24}$  and  $AUC_{0-\infty}$ . PK parameters will be determined using noncompartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, SD, coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

For calculation of mean concentrations and generation of mean concentration-time profiles, all below the limit of quantification (BLQ) values will be set to zero except when an individual BLQ falls between 2 quantifiable values, in which case it will be omitted.

If there are values above the BLQ, but too sparse to allow full analysis, descriptive statistics will be performed on available values.

Syntimmune, Inc.  Final 18 January 2017

#### 12.5 Safety Data

Safety observations and measurements include AEs, safety laboratory tests, vital sign measurements, PEs, and ECGs.

Treatment-emergent AEs will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

AEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject, cohort, and overall per SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by cohort. Incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the local laboratory.

Vital sign measurements and change from baseline will be summarized at each scheduled time point by cohort using descriptive statistics.

Arithmetic mean of parameters from triplicate ECG will be calculated first for each participant at each planned time point. Then summary statistics of ECG test parameters (mean of triplicate) and change from baseline to each post-dose time point will be calculated. Shift tables for ECG test result category change (normal, abnormal, clinically abnormal) from pre-dose to each post-dose time point showing number and percentage of subjects with movement between categories will be presented by treatment group. Frequency and percentage of subjects experiencing potential QTc prolongation (QTcF > 450) will be summarized at each time point by cohort.

#### 12.6 Pharmacodynamic/Activity Data

PD results will be summarized by cohort.

#### 12.7 Immunogenicity Data

Immunogenicity results will be summarized by cohort.

## 12.8 Interim Analysis

No interim analysis is planned. Safety results will be examined for making dose-escalation decisions; no statistical analyses are planned for aiding these dose-escalation decisions.

#### 13 DATA QUALITY ASSURANCE

All data will be entered in a validated electronic data capture system using single data entry. Standard procedures (including following data review guidelines, manual clinical review based on subject profiles, computerized validation to produce queries, and maintenance of an audit file which includes all database modifications) will be followed to ensure accurate data. Clinical personnel will review all data listings for outliers, data inconsistencies, and spelling errors.

During the study, a study site monitor will make site visits to review protocol compliance, compare electronic case report forms (eCRFs) against individual subject medical records, assess drug accountability, and ensure that the study is being conducted using pertinent regulatory requirements. eCRF entries will be verified with source documentation. The review of medical records will be performed in a manner to ensure that subject confidentiality is maintained. Checking the eCRFs for completeness, clarity and cross checking with source documents is required to monitor the progress of the study. Direct access to source data is also required for inspections and audits, and will be carried out giving due consideration to data protection and medical confidentiality. Each Investigator will have assured Syntimmune of full access to complete source data for study participants and associated necessary support at all times.

In addition to routine monitoring procedures, audits of clinical research activities in accordance with standard operating procedures (SOPs) may be performed to evaluate compliance with the principles of GCP. A regulatory authority may also wish to conduct an inspection (during the study or even after its completion). If a regulatory authority requests an inspection, the Investigator must immediately inform Syntimmune that this request has been made. Study conduct may be assessed during the study by a Clinical Quality Assurance representative(s) to ensure that the study is conducted in compliance with the protocol. This designee, as well as the site monitor, will be permitted to inspect the study documents (study protocol, eCRFs, investigational product accountability, original study-relevant medical records). All subject data will be treated confidentially. During the clinical study, access will be available to Syntimmune or their designee (e.g., contract research organization [CRO]) to view the eCRFs after completion of the individual sections of the study. Furthermore, the study protocol, each step of the data-recording procedure and the handling of the data as well as the study report may be subject to independent review by a Quality Assurance representative. Clinical site and study audits will be conducted as necessary to assure the validity of the study data.

#### 14 STUDY ADMINISTRATION

#### 14.1 Study Administrative Structure

The study administration structure is provided in Table 6.

**Table 6:** Study Administrative Structure



#### 14.2 Ethical Conduct of the Study

The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH E6 Tripartite Guideline (January 1997), and in general, be conducted in a manner consistent with the principles described in the Declaration of Helsinki. The Investigator will ensure that the conduct of the study complies with the basic principles of GCP as outlined in the current version of 21 CFR, subpart D, Part 312, "Responsibilities of Sponsors and Investigators", Part 50, "Protection of Human Subjects", and Part 56, "Institutional Review Boards".

#### 14.3 Informed Consent (ICF)

A properly executed, written informed consent document, in compliance with 21 CFR, Part 50 and the ICH guidelines, will be obtained from each subject before the subject is entered into the study and before any study screening procedure is performed that involves risk. Attention will

Syntimmune, Inc.  Final 18 January 2017

be directed to the basic elements required for incorporation into the informed consent under US Federal Regulations for Protection of Human Subjects (21 CFR 50.25[a]) and (21 CFR 50.25[b]), as necessary.

Sample ICFs will be supplied to each site. Syntimmune or its designee must review any proposed deviations from the sample ICF. The final IRB-approved document must be provided to Syntimmune for regulatory purposes.

It is the responsibility of the Investigator, or a person designated by the Investigator, to obtain written informed consent from each subject (or the subject's legally authorized representative) participating in this study after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study. In the case where the subject is unable to read, an impartial witness should be present during the entire informed consent discussion. After the subject has orally consented to participation in the trial, the witness' signature on the form will attest that the information in the consent form was accurately explained and understood. A copy of the ICF must be provided to the subject or to the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

The eCRF for this study contains a section for documenting informed subject consent, and this must be completed appropriately. Signed ICFs must remain in each subject's study file and must be available for verification by site monitors at any time. If new safety information results in significant changes in the risk/benefit assessment, the consent form should be reviewed and updated as necessary. All subjects (including those already being treated) should be informed of the new information, should be given a copy of the revised form, and should give their consent to continue in the study.

#### 14.4 Institutional Review Board

This study is being conducted under US IND 128152. This protocol (and any modifications) and appropriate consent procedures must be reviewed and approved by an IRB. This board must operate in accordance with the current federal or local regulations. The Investigator will send a letter or certificate of IRB approval to Syntimmune (or designee) before subject enrollment and whenever subsequent modifications to the protocol are made.

#### **14.5 Dose Escalation Committee**

The DEC will be responsible for confirming the safety of the investigative product prior to dose escalation, as well as the dose level for each successive cohort. In addition, over the course

Syntimmune, Inc.  Final 18 January 2017

of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects. The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions.

#### 14.6 Future Use of Subject Samples

Not all the tissue and blood components obtained during this study may be required for the tests that are part of the clinical trial. Available samples may be used for additional research. This research will help to understand disease subtypes, drug response and AE, and possibly identify new drug targets or biomarkers that predict subject response to treatment. The use of the samples for internal research will be done using the guidelines defined by the FDA guidance for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individual Identifiable (issued 25 April 2006) and the European Medicines Agency (EMA) Reflection Paper on Pharmacogenetic Samples, Testing and Data Handling (Doc. Ref.

EMEA/CHMP/PGxWP/201914/2006; 15 November 2007). If a subject requests destruction of their tissue and blood samples and the samples have not yet been de-identified, Syntimmune will destroy the samples as described in this FDA guidance. Syntimmune will notify the Investigator in writing that the samples have been destroyed.

#### 15 CONDITIONS FOR MODIFYING THE PROTOCOL

Protocol modifications to ongoing studies must be made only after consultation between a Syntimmune representative and the Investigator. Protocol modifications will be prepared, reviewed, and approved by Syntimmune representatives.

All protocol modifications must be submitted to the IRB for information and approval in accordance with local requirements, and to regulatory agencies if required. Approval must be obtained before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to study subjects, or when the change involves only logistical or administrative aspects of the trial (e.g., change in site monitor, change of telephone number).

#### 16 CONDITIONS FOR TERMINATING THE STUDY

Syntimmune has the right to terminate the study at any time. In terminating the study, Syntimmune and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests.

#### 17 STUDY DOCUMENTATION, CRFS, AND RECORD KEEPING

#### 17.1 Investigator's Files and Retention of Documents

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into 2 separate categories as follows: (1) Investigator's study file and (2) subject clinical source documents.

The Investigator's study file will contain the protocol and protocol amendments, eCRFs, query forms, IRB and governmental approval with correspondence, sample informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

Subject clinical source documents (usually predefined by the project to record key efficacy and safety parameters independent of the eCRFs) may include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, electroencephalogram, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject screening and enrollment logs. The Investigator must keep these 2 categories of documents on file for at least 2 years following the marketing application approval date for the study treatment and for the indication being investigated or for 2 years after the development program is discontinued and the FDA notified. After that period, the documents may be destroyed subject to local regulations with prior written permission from Syntimmune. If the Investigator wants to assign the study records to another party or move them to another location, Syntimmune must be notified in advance.

If the Investigator cannot guarantee the archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and Syntimmune to store these in a sealed container outside of the study site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storing outside of the study site.

#### 17.2 Source Documents and Background Data

Investigators must maintain adequate and accurate source documents on which the eCRFs for each subject are based. They are separate and distinct from the eCRFs.

These records include detailed notes on the following:

- Medical history
- Date and time of informed consent with Health Insurance Portability and Accountability
  Act (HIPAA) authorization either contained in the ICF or presented to the subject
  candidate as a standalone document
- Description of the complete consenting process
- The basic identifying information that linked the subject's medical record with the eCRFs
- The results of all diagnostic tests performed, diagnoses made, therapy provided, and any other data on the condition of the subject
- The medical condition of the subject during their involvement in the study
- All AEs
- The subject's exposure to the study medication
- The subject's exposure to any concomitant therapy
- All relevant observations and data on the condition of the subject throughout the trial
- Justification for all entries in the subject's eCRF

A subject log of all potentially eligible subjects considered, but not consented, for obvious deviations from the entry criteria, will be kept at each site. The log will contain subjects' initials, diagnosis, eligibility, or, if not eligible, reason for not consenting. All consented subjects will be logged, regardless of whether they ultimately enroll.

Upon request, the Investigator will supply Syntimmune with any required background data from the study documentation or clinic records. This is particularly important when eCRFs are illegible or when errors in data transcription are suspected. In case of special problems or governmental queries or requests for audit inspections, it is also necessary to have access to the complete study records, provided that subject confidentiality is protected.

#### 17.3 Audits and Inspections

The Investigator should understand that source documents for this study should be made available to appropriately qualified personnel from Syntimmune (or designee), or to health authority inspectors after appropriate notification. The verification of the eCRF data must be by direct inspection of source documents.

#### 17.4 Electronic Case Report Forms

Clinical trial data for this study will be captured on eCRF designed for computer processing and analysis. This computerized system will be validated and compliant with 21 CFR Part 11. Corrections to data will be made using 21 CFR Part 11, Electronic Records; Electronic Signatures. If corrections are made after review and sign-off by the Investigator, he/she must be aware of the changes and provide written acknowledgement. There will also be an electronic audit trail. Corrections on paper CRFs must be initialed and dated by the person making the change. The Investigator agrees to provide all information requested on the eCRF in an accurate manner using instructions provided. The Investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported to Syntimmune in the eCRF and in all required reports.

An eCRF is required to be submitted for every subject who receives any amount of study drug. This includes submission of retrievable data on subjects who withdraw before completion of the study. Prior to submission, eCRFs must be reviewed for completeness and accuracy, and signed and dated where either indicated, by the Principal Investigator or authorized delegate from the study staff. If a subject stops treatment or terminates from the study, the dates and reasons must be noted on the eCRF.

#### 18 MONITORING THE STUDY

It is understood that the responsible Syntimmune site monitor (or designee) will contact and visit the Investigator regularly and will be allowed on request to inspect the various records of the trial (eCRFs and other pertinent data) if subject confidentiality is maintained in accordance with local requirements.

It will be the site monitor's responsibility to inspect the eCRFs at regular intervals throughout the study, to verify the adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The site monitor should have access to laboratory test reports and other subject records needed to verify the entries on the eCRF. The Investigator (or designee) must agree to cooperate with the site monitor to ensure that any problems detected during these monitoring visits are resolved.

#### 19 CONFIDENTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECORDS

The Investigator must ensure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On eCRFs or other documents submitted to Syntimmune, subjects should be identified by an identification code and not by their names. The Investigator should keep a subject enrollment log showing codes, names, and addresses. The Investigator should maintain documents not for submission to Syntimmune (e.g., subjects' written consent forms) in strict confidence.

Authorized regulatory officials and Syntimmune personnel (or their representatives) will be allowed full access to inspect and copy the records. All study drugs, subject bodily fluids and tissue, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by Syntimmune.

The Principal Investigator also agrees that all information received from Syntimmune, including but not limited to the IB, this protocol, eCRFs, the INDs, and any other study information remain the sole and exclusive property of Syntimmune during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from the sponsor. The Principal Investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 20 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. The Investigator agrees that any manuscript or abstract they author may be published only after receiving written permission from Syntimmune.

If Syntimmune coordinates a publication or presentation of study results from all study sites, the participation of Investigator or other representatives of study site as a named author shall be determined in accordance with Syntimmune policy and generally accepted standards for authorship.

#### 21 REFERENCES

Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID), which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. *Clin. Exp. Immunol.* 2013;174: 203-211.

Bugelski PJ and Treacy G. (2004) Predictive power of preclinical studies in animals for the immunogenicity of recombinant therapeutic proteins in humans. *Curr Opin Mol Ther*. 2004;6:10–16.

International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) (2011). S6(R1) Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals. Accessed 03 June 2016.

http://www.ich.org/products/guidelines/safety/safety-single/article/preclinical-safety-evaluation-of-biotechnology-derived-pharmaceuticals.html

Nixon AE, Chen J, Sexton DJ, Muruganandam A, Bitonti AJ, Dumont J, Viswanathan M, Martik D, Wassaf D, Mezo A, Wood CR, Biedenkapp JC, TenHoor C. (2015). Fully human monoclonal antibody inhibitors of the neonatal Fc receptor reduce circulating IgG in non-human primates. Front. Immun. 6:176

Ponce R, Abad L, Amaravadi, L, et al. Immunogenicity of biologically-derived therapeutics: assessment and interpretation of nonclinical safety studies. *Regul Toxicol Pharmacol*. 2009;54,164–182.

Roopenian, D.C., Christianson, G.J., Sproule, T.J., Brown, A.C., Akilesh, S., Jung, N., Petkova, S., Avanessian, L., Choi, E.Y., Shaffer, D.J., Eden, P.A., Anderson, C. L. The MHC class I-like IgG receptor controls perinatal IgG transport, IgG homeostasis, and fate of IgG-Fc-coupled drugs. 2003. J. Immun. 170 3528-3533

Appendix A: NCI CTCAE, Version 4.03

# Common Terminology Criteria for Adverse Events (CTCAE)

## Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

#### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

### Common Terminology Criteria for Adverse Events v4.0 (CTCAE) Publish Date: May 28, 2009

#### Quick Deference

The NCI Common Terminology Criteria for A brief definition is provided Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

#### **Components and Organization**

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### CTCAE Terms

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest A Semi-colon indicates 'or' within the description Level Term).

#### Definitions

to clarify the meaning of each AE term.

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical and therefore is not an option. descriptions of severity for each AE based on this general guideline:

Grade 1 Mild: asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not

noninvasive intervention indicated; limiting age-appropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.

Life-threatening Grade 4 consequences: urgent intervention indicated.

Grade 5 Death related to AE.

of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs

#### Activities of Daily Living (ADL)

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

\*\*Self care ADL refer to bathing, dressing and Grade 2 Moderate; minimal, local or undressing, feeding self, using the toilet, taking medications, and not bedridden.

<sup>+</sup> CTCAE v4.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).

#### CONTENTS

| SOC | Page |
|---------------------------------------------------------------------|------|
| Blood and lymphatic system disorders | 3 |
| Cardiac disorders | 4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 9 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | 76 |
| Vascular disorders | 77 |

| Blood and lymphatic system disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Anemia | Hemoglobin (Hgb) <lln -="" 10.0<br="">g/dL; <lln -="" -<br="" 6.2="" <lln="" l;="" mmol="">100 g/L</lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an reduction in the amount of palpitations of the heart, soft syst | • | • • • | ay include pallor of the skin and m | iucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25% reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50% reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder characteriz | ed by the inability of the bone mar | row to produce hematopoietic ele | ments. | | |
| Disseminated intravascular<br>coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by systemic pathological activa<br>s depleted of platelets and coagula | - | which results in clot formation thro | oughout the body. There is an incr | ease in the |
| Febrile neutropenia | - | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>degrees F) for more than one ho | ed by an ANC <1000/mm3 and a sur. | single temperature of >38.3 degre | es C (101 degrees F) or a sustaine | ed temperature of >=38 degrees 0 | (100.4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate widespread erythrocyte ce | Il membrane destruction. | I | |
| Hemolytic uremic syndrome | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteriz | ed by a form of thrombotic microa | ngiopathy with renal failure, hemo | lytic anemia, and severe thromboo | ytopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of leucostasis; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate an increased number of w | nite blood cells in the blood. | | |
| Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in a lymph node. | | | |
| Spleen disorder | Incidental findings (e.g., Howell-<br>Jolly bodies); mild degree of<br>thrombocytosis and<br>leukocytosis | Prophylactic antibiotics indicated | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder of the splee | en. | | | | |
| Thrombotic thrombocytopenic<br>purpura | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | ed by the presence of microangion al disturbances. It is an acute or s | • | cytopenic purpura, fever, renal abr | normalities and neurological abnor | malities suc |
| Blood and lymphatic system | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| disorders - Other, specify | symptoms; clinical or diagnostic observations only; intervention not indicated | noninvasive intervention indicated; limiting age-appropriate instrumental ADL | but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | urgent intervention indicated | |

| Cardiac disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute coronary syndrome | - | Symptomatic, progressive angina; cardiac enzymes normal; hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | | • | dium secondary to coronary artery | disease. The clinical presentation | covers a |
| | unstable angina to myocardial infa | | I | | I |
| Aortic valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in aortic valve func | tion or structure. | I | I | 1 |
| Asystole | Periods of asystole; non-urgent medical management indicated | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia without cardi | ac electrical activity. Typically, this | is accompanied by cessation of the | ne pumping function of the heart. | |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>originates above the ventricles. | ed by a dysrhythmia without disce | rnible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz atria. | ed by a dysrhythmia with organize | ed rhythmic atrial contractions with | a rate of 200-300 beats per minut | e. The rhythm disturbance origina | tes in the |
| Atrioventricular block complete | - | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with complete | e failure of atrial electrical impulse | conduction through the AV node t | to the ventricles. | |
| Atrioventricular block first<br>degree | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | - | - | - |
| | ed by a dysrhythmia with a delay interval greater than 200 milliseco | • | tion of an electrical impulse throug | gh the atrioventricular (AV) node b | eyond 0. |
| Cardiac arrest | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by cessation of the pumping fu | nction of the heart. | | | |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by substernal discomfort due to | insufficient myocardial oxygenati | on. | | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by pathological irregularities in | the cardiac conduction system. | 1 | | , |
| Constrictive pericarditis | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | 1 | ı | 1 . | 1 | e action. |
| Definition: A disorder characteriz | ed by a thickened and fibrotic peri | cardial sac; these fibrotic changes | impede normal myocardiai functio | | |

| Cardiac disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic<br>dysfunction | - | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | zed by failure of the left ventricle to<br>nea, orthopnea, and other signs ar | | e an increase in distending pressur<br>stion and edema. | e and in end-diastolic volume. Clin | ical |
| Mitral valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | zed by a defect in mitral valve func | tion or structure. | | | 1 |
| Mobitz (type) II atrioventricular<br>olock | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a dysrhythmia with relatively<br>atrioventricular (AV) node to the ve | • | block of an atrial impulse. This is t | he result of intermittent failure of a | trial elect |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a progre<br>on through the atrioventricular (AV | | rior to the blocking of an atrial impu | alse. This is the result of intermitter | nt failure o |
| Myocardial infarction | - | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences;<br>hemodynamically unstable | Death |
| Definition: A disorder characteriz | red by gross necrosis of the myoca | ardium; this is due to an interruption | on of blood supply to the area. | | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or<br>with minimal activity or exertion;<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characteriz | red by inflammation of the muscle | tissue of the heart. | | 1 | |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | - | - | - |
| Definition: A disorder characterize | red by an unpleasant sensation of | irregular and/or forceful beating o | f the heart. | T | 1 |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characteriz<br>originates in the atria. | red by a dysrhythmia with abrupt o | nset and sudden termination of at | trial contractions with a rate of 150- | -250 beats per minute. The rhythm | disturba |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by fluid collection within the pe | ricardial sac, usually due to inflam | nmation. | | |
| Pericardial tamponade | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| | rad by an increase in intrancricardi | al pressure due to the collection of | of blood or fluid in the pericardium. | | |
| Definition: A disorder characteriz | eu by an increase in intrapencardi | | | | |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in pulmonary valve | function or structure. | i | i | |
| Restrictive cardiomyopathy | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | ted by an inability of the ventricles | | | | I |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., ventricular assist device);<br>heart transplant indicated | Death |
| Definition: A disorder characteriz | ed by impairment of right ventricul | ar function associated with low eje | ection fraction and a decrease in n | notility of the right ventricular wall. | |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with alternation | | | | |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical intervention indicated | Severe, medically significant, medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate less than 60 beats per minute | that originates in the sinus node. | | |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates in the sinus no | ode. | |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates above the ven | tricles. | 1 |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| | ed by a defect in tricuspid valve fu | | | I | I |
| Ventricular arrhythmia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by a dysrhythmia that originate | s in the ventricles. | I | 1 | 1 |
| Ventricular fibrillation | - | - | - | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz ventricles. | ed by a dysrhythmia without disce | rnible QRS complexes due to rapi | d repetitive excitation of myocardi | al fibers without coordinated contr | action of the |
| Ventricular tachycardia | - | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates distal to the bu | undle of His. | |
| Wolff-Parkinson-White<br>syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of an accessor | ry conductive pathway between th | e atria and the ventricles that caus | ses premature ventricular activatio | n. |
| Cardiac disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Congenital, familial and genetic disorders | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Congenital, familial and genetic | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| disorders - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| i | | | disabling; limiting self care ADL | | |

| Ear and labyrinth disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | mfort in the ear. | | | |
| External ear inflammation | External otitis with erythema or dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis;<br>stenosis or osteomyelitis;<br>necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation, swelling and r | edness to the outer ear and ear c | anal. | • | , |
| External ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | mfort in the external ear region. | | • | |
| Hearing impaired | Adults enrolled on a Monitoring<br>Program (on a 1, 2, 3, 4, 6 and<br>8 kHz audiogram): Threshold<br>shift of 15 - 25 dB averaged at 2 | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 4 kHz and above in at least one ear. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated. Adults not enrolled in Monitoring Program: hearing loss with hearing aid or intervention indicated; limiting self care ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids; threshold shift >20 dB at 3 kHz and above in at least one ear; additional speech-language related services indicated. | Adults: Decrease in hearing to profound bilateral loss (absolute threshold >80 dB HL at 2 kHz and above); non-servicable hearing. Pediatric: Audiologic indication for cochlear implant and additional speech-language related services indicated. | - |
| Definition: A disorder characte | ा<br>rized by partial or complete loss of th | ।<br>le ability to detect or understand s | 1 | ı<br>ar structures. | ı |
| Middle ear inflammation | Serous otitis rized by inflammation (physiologic re | Serous otitis, medical intervention indicated | Mastoiditis; necrosis of canal soft tissue or bone | Life-threatening consequences; urgent intervention indicated | Death |
| Finnitus | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by noise in the ears, such as ri | nging, buzzing, roaring or clicking. | Г | Г | |
| /ertigo | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte<br>vertigo). | rized by a sensation as if the externa | ll world were revolving around the | patient (objective vertigo) or as if | he himself were revolving in space | e (subjectiv |
| Vestibular disorder | - | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by dizziness, imbalance, nause | a, and vision problems. | | | |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Endocrine disorders | | | | | | | |
|---|---|---|---|---|---|--|--|
| | | | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 | | |
| Adrenal insufficiency | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death | | |
| | urs when the adrenal cortex does not<br>dison's disease or primary adrenal ins | | cortisol and in some cases, the ho | rmone aldosterone. It may be due | to a disord | | |
| Cushingoid | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms, medical intervention or hospitalization indicated | - | - | | |
| Definition: A disorder characte<br>osteoporosis, usually due to e | erized by signs and symptoms that re<br>xogenous corticosteroids. | semble Cushing's disease or synd | drome: buffalo hump obesity, striat | ions, adiposity, hypertension, diab | etes, and | | |
| Delayed puberty | - | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | - | - | | |
| Definition: A disorder characte | rized by unusually late sexual maturi | ty. | | | | | |
| Growth accelerated | - | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | - | - | | |
| Definition: A disorder characte | erized by greater growth than expecte | d for age. | 1 | | | | |
| Hyperparathyroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - | | |
| Definition: A disorder characte the blood). | rized by an increase in production of | parathyroid hormone by the para | thyroid glands. This results in hype | ercalcemia (abnormally high levels | of calcium | | |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid suppression therapy indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death | | |
| Definition: A disorder characte | erized by excessive levels of thyroid h | ormone in the body. Common car | uses include an overactive thyroid | gland or thyroid hormone overdos | ie. | | |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical intervention or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death | | |
| Definition: A disorder characte | rized by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | | | | |
| Hypothyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death | | |
| | erized by a decrease in production of | | and. | 1 | | | |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical<br>markers of puberty for females<br><8 years and males <9 years | - | | - | | |
| Definition: A disorder characte<br>9 for boys. | erized by unusually early developmen | t of secondary sexual features; th | e onset of sexual maturation begin | ns usually before age 8 for girls an | d before ag | | |
| Virilization | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - | | |
| Definition: A disorder characte | rized by inappropriate masculinization | n occurring in a female or prepub | ertal male. | <del>,</del> | | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death | | |
| Intervention indicated (e.g., topical agents); limiting soft care (20/200 or worse) in the affected eye and an afterior chamber. By a symptomatic; clinical or diagnostic observations only instrumental ADL affected eye affected eye affected eye and an affect of the comea. It is associated with inflammatory cells in the comea and anterior chamber. By a symptomatic; clinical or diagnostic observations only instrumental ADL affected eye affected e | | | Eye dis | sorders | | |
|---|---|---|---|---|---|---|
| Ellured vision Intervention not indicated Symptomatic, initiality Cambridge performance of ADL - | | | | Grade | | |
| Definition: A disorder characterized by visual perception of trustees or thizy images. Cational Asymptomatic, clinical or disoption of trustees or thizy images. Cational Asymptomatic, clinical or disoption of trustees or thizy images. Cational Asymptomatic, clinical or disoption of trustees or thizy images. Corp. Asymptomatic moderated by partial or complete opecity of the crystalline lens of one or both eyes. This results in a decrease in visual actually and eventual blinchess of underlined and included or disoptions. Intervention industed by inflammation, swelling architecture of the eye. Corp. Corp. Asymptomatic moderated by inflammation, swelling architecture, included or disoptions intervention industed by an area of aphthetis trustees or the corp. Symptomatic, metical algorithms of the eye. Corp. Corp. Asymptomatic clinical or disoptions of the eye or disoptions or the eye or disoptions or the eye or disoptions or the eye or disoptions or the eye or disoptions. Intervention industed by an area of aphthetis trustees or the corp. Asymptomatic clinical or disoptions or the eye or disoptions or t | Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Apyrophomatic: directary of agreements conservations only intervention and indicated or agreement for conservation (apyrophomatic) and conservation (apyrophomatic) a | | | instrumental ADL | Limiting self care ADL | - | - |
| diagnostic cherevation on processes in visual acuity of the effective dependence of the content of the affected services and acuity of the content of the co | | 1 | 1 | I | | |
| Definition: A disorder characterized by partial or complete opacity of the crystalline lens of one or both eyes. This results in a decrease in visual acuity and eventual blindness if untiversition. Asymptoms: intervention indicated (e.g., supplementations) in the viterous humanor or lens. Elevated intervention indicated (e.g., supplementation indicated (e.g., su | Cataract | diagnostic observations only; | decrease in visual acuity | decrease in visual acuity<br>(worse than 20/40 but better<br>than 20/200); operative<br>intervention indicated (e.g., | , | - |
| Asymptomatic or mild symptoms intervention on indicated by inflammation, average and intervention indicated (e.g., ariselected by inflammation, average and indicated (e.g., ariselected by inflammation, average and indicated (e.g., ariselected by inflammation, average and indicated (e.g., ariselected by an area of epithelial tissue loss on the surface of the company store of the eye. Definition: A disorder characterized by an area of epithelial tissue loss on the surface of the comea. It is associated with inflammatory cells in the cornea and anterior chamber. | | ।<br>erized by partial or complete op | i<br>eacity of the crystalline lens of c | | ।<br>। a decrease in visual acuity ar | I<br>nd eventual blindness if |
| Comeal ulder | | symptoms; intervention not | intervention indicated (e.g., antibiotics); limiting | Limiting self care ADL | - | - |
| Intervention indicated (e.g., topical agents); limiting instrumental ADL Intervention indicated (e.g., topical agents); limiting instrumental ADL Intervention indicated (e.g., topical agents) in the cornea and anterior chamber. | Definition: A disorder characte | erized by inflammation, swelling | and redness to the conjunctiv | a of the eye. | | |
| Dry eye Asymptomatic; clinical or diagnostic observations only; mild symptoms relieved by Unbricants Definition: A disorder characterized by dryness of the cornea and conjunctiva. Extraocular muscle paresis Asymptomatic; clinical or diagnostic observations only Instrumental ADL Instrumenta | Corneal ulcer | - | intervention indicated (e.g., topical agents); limiting | declining vision (worse than | (20/200 or worse) in the | - |
| diagnostic observations only, mild symptoms relieved by lubricants Definition: A disorder characterized by dynness of the comes and conjunctiva. Extracoular muscle paresis Asymptomatic, clinical or diagnostic observations only instrumental ADL Limiting self care ADL; disabiling - | Definition: A disorder characte | erized by an area of epithelial ti | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the cornea | and anterior chamber. |
| Extraocular muscle paresis | Dry eye | diagnostic observations only;<br>mild symptoms relieved by | agents indicated; limiting | (<20/40); limiting self care | - | - |
| Definition: A disorder characterized by incomplete paralysis of an extraocular muscle. Eye pain Mild pain Moderate pain; limiting self care ADL care ADL care ADL: Symptomatic; clinical or diagnostic observations only intervention not indicated intervention in clinicated: Symptomatic but not limiting ADL Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only intervention not indicated intervention indicated: Initial parameterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Eliovated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficits (e.g., involving topical agent for intervention; no visual field deficit. In visual field deficit. Symptomatic but not limiting and the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting agents, limiting agent care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting agents, limiting instrumental ADL Definition: A disorder characterized by an increase in pressure of the eye. Night blindness Symptomatic but not limiting ADL Limiting self care ADL - a service and the care add the ca | Definition: A disorder characte | erized by dryness of the cornea | and conjunctiva. | | | |
| Eye pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated of limiting instrumental ADL intervention indicated; limiting instrumental ADL perintion: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Elimiting instrumental ADL and part of light. Floaters Symptomatic but not limiting Limiting instrumental ADL ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit; multiple topical or or al agents indicated; limiting instrumental ADL with ging instrumental ADL with ging instrumental ADL. Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic indicated (e.g., involving self care ADL in the affected eye of the previous of the aqueous humor outflow. Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL blimiting sel | Extraocular muscle paresis | | | | - | - |
| Instrumental ADL Care ADL | Definition: A disorder characte | erized by incomplete paralysis | of an extraocular muscle. | | | |
| Eyelid function disorder diagnostic observations only; intervention indicated: intervention indicated; limiting self care ADL; operative intervention indicated: poperative intervention poperative intervention poperati | Eye pain | Mild pain | | | - | - |
| diagnostic observations only; intervention indicated; limiting instrumental ADL initing instrumental ADL initing instrumental ADL initing self care ADL - | Definition: A disorder characte | erized by a sensation of marked | d discomfort in the eye. | T | | 1 |
| Flashing lights Symptomatic but not limiting ADL ADL Limiting instrumental ADL ADL Limiting self care ADL | Eyelid function disorder | diagnostic observations only; | intervention indicated; | operative intervention | - | - |
| Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit limiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL ElOP causing marked visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Declinition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) and intervention in the vitreous humor or lens. ElOP causing marked visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Blindness (20/200 or worse) in the affected eye - | | | | I | | 1 |
| Symptomatic but not limiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting ADL Continuiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting ADL Limiting self care ADL Continuiting Self care ADL Continuiting ADL Limiting self care ADL Limiting self care ADL Continuiting Self care ADL Continuiting Self care ADL Continuiting ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL Continuiting Self care ADL | Flashing lights | | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Elevated intraocular pressure (ElOP) with single topical agent for intervention; no visual field deficits; multiple topical or oral agents indicated; limiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents; limiting agents; limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Blindness (20/200 or worse) in the affected eye - Limiting self care ADL Blindness (20/200 or worse) in the affected eye - Limiting self care ADL Blindness (20/200 or worse) in the affected eye - Limiting self care ADL Blindness (20/200 or worse) in the affected eye - Limiting self care ADL Blindness (20/200 or worse) in the affected eye | Definition: A disorder characte | erized by a sudden or brief burs | st of light. | I | | T |
| Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit (limiting instrumental ADL pefinition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL pefinition: A disorder characterized by inflammation to the cornea of the eye. EIOP causing marked visual field deficits (e.g., involving both superior and inferior visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL and affected eye Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) in the affected eye - In the affected eye - In the affected eye - In the affected eye | Floaters | | Limiting instrumental ADL | Limiting self care ADL | - | - |
| pressure (EIOP) with single topical agent for intervention; no visual field deficit Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting ADL Limiting instrumental ADL Itimiting self care ADL | Definition: A disorder characte | erized by an individual seeing s<br>T | pots before their eyes. The sport | ots are shadows of opaque cell | fragments in the vitreous hum | or or lens. |
| Keratitis - Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL Decline in vision (worse than 20/200 or worse) in the affected eye (20/200 or worse) in the affected eye Limiting self care ADL Blindness (20/200 or worse) in the affected eye - In the affected eye | Glaucoma | pressure (EIOP) with single topical agent for intervention; | field deficits; multiple topical or oral agents indicated; | field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated; | · ' | - |
| intervention indicated (e.g., topical agents); limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Blindness (20/200 or worse) in the affected eye Limiting self care ADL in the affected eye | Definition: A disorder characte | erized by an increase in pressu | re in the eyeball due to obstruc | tion of the aqueous humor out | low. | |
| Night blindness Symptomatic but not limiting ADL Limiting self care ADL Blindness (20/200 or worse) - in the affected eye | | - | intervention indicated (e.g., topical agents); limiting instrumental ADL | 20/40 but better than 20/200); limiting self care | (20/200 or worse) in the | - |
| ADL in the affected eye | Definition: A disorder characte | | ornea of the eye. | T | | 1 |
| | Night blindness | | Limiting instrumental ADL | Limiting self care ADL | , | - |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only | Limiting vision of the affected eye (20/40 or better) | eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| | erized by involvement of the op | · | i | | 1 |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by swelling around the o | ptic disc.<br>T | <u> </u> | <u> </u> | |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charact | erized by fear and avoidance of | f light. | | | |
| Retinal detachment | Asymptomatic | Exudative and visual acuity<br>20/40 or better | Rhegmatogenous or<br>exudative detachment;<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by the separation of the | inner retina layers from the und | derlying pigment epithelium. | | |
| Retinal tear | - | Laser therapy or pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by a small laceration of t | he retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | s and floaters. |
| Retinal vascular disorder | - | Topical medication indicated | Intravitreal medication; operative intervention indicated | - | - |
| Definition: A disorder charact | erized by pathological retinal bl | ood vessels that adversely affe | ects vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked<br>decrease in visual acuity<br>(worse than 20/40);<br>disabling; limiting self care<br>ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder involvin | g the retina. | | | | |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better) | Symptomatic, limiting self care ADL; marked decrease in visual acuity (worse than 20/40) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by involvement of the so | lera of the eye. | T | Τ | I |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | • | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by inflammation to the uv | vea of the eye. | ı | i - | 1 |
| Vitreous hemorrhage | Asymptomatic or mild symptoms; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by blood extravasation in | nto the vitreous humor. | T | T | T |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | - | - |
| Definition: A disorder of excess | ssive tearing in the eyes; it can | be caused by overproduction of | of tears or impaired drainage of | the tear duct. | |
| Eye disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care | Sight-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by swelling of the abdomen. | | | | 1 |
| Abdominal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the abdominal region. | T | | 1 |
| Anal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the opening in the anal | canal to the perianal skin. | | |
| Anal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the anal region | on. | T | | 1 |
| Anal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the mucous | membrane of the anus. | ı | | |
| Anal necrosis | - | - in the engl region | TPN or hospitalization indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by a necrotic process occurring | | Cavara naint limiting calf care | | |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | erized by a sensation of marked disco | | 0 1 1 1 | Let up a control of the control of t | <b>.</b> |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the anal canal. | | | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the anal ca | nal. | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by accumulation of serous or h | emorrhagic fluid in the peritoneal | cavity. | • | |
| Bloating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | - | - | - |
| Definition: A disorder characte | erized by subject-reported feeling of u | incomfortable fullness of the abdo | men. | | |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the cecum. | | | | |
| Cheilitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | - | - |
| | | I | I | I | I . |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| Advance France | | | Grade | | Ι, |
| Adverse Event | 1 | 2 | 3 | 4 | |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the colon. | | | | |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the large intestine and | another organ or anatomic site. | | |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the colon. | T | T | Γ | |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated rized by blockage of the normal flow | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | Tized by blockage of the normal flow | | | | D41- |
| Colonic perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by a rupture in the colonic wall. | | | | 1 |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the colon. | ' | ' | • |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the colon. | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with regular use of laxatives or enemas; limiting instrumental ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by irregular and infrequent or d | ifficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis or periapical abscess or resulting in tooth loss | - | - |
| Definition: A disorder characte | rized by the decay of a tooth, in whice | h it becomes softened, discolored | and/or porous. | | |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day over baseline; moderate increase in ostomy output compared to baseline | Increase of >=7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by frequent and watery bowel n | novements. | | | |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment orally; tube feeding or TPN indicated; unstimulated saliva <0.1 ml/min | - | - |

| | | Gastrointestinal disorders | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the duodenum and and | other organ or anatomic site. | | |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the duodenur | n. | | | |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective operative intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of stomach contents through the | duodenum. | | |
| Duodenal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a rupture in the duodenal w | all. | T | 1 | 1 |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the duodenum. | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the duoder | nal wall. | |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | erized by an uncomfortable, often pai | nful feeling in the stomach, resulti | ing from impaired digestion. Sympt | oms include burning stomach, blo | ating, |
| heartburn, nausea and vomiti | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely altered eating/swallowing; tube feeding or TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by difficulty in swallowing. | 1 | | ı | 1 |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent abdominal pain; fever; ileus; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the small ar | nd large intestines. | _ | | |
| Enterovesical fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the urinary bladder and | d the intestine. | | |
| Esophageal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the esophagus and and | other organ or anatomic site. | | |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |

| Gastrointestinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | g in the esophageal wall. | | | |
| Esophageal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by blockage of the normal flow | | | | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the esophageal region. | | | |
| Esophageal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a rupture in the wall of the e | 1 | | 1 | |
| Esophageal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the esophagus. | | <b>.</b> | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammate | ory and necrotic erosive lesion on | the mucosal surface of the esopha | geal wall. | |
| Esophageal varices<br>hemorrhage | - | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from esophageal v | arices. | | | |
| Esophagitis Definition: A disorder characte | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered eating/swallowing; oral supplements indicated | Severely altered<br>eating/swallowing; tube feeding,<br>TPN or hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Fecal incontinence | Occasional use of pads required | | Severe symptoms; elective | - | - |
| | | | operative intervention indicated | | |
| Definition: A disorder characte | rized by inability to control the escap | e of stool from the rectum. | | T | |
| Flatulence | Mild symptoms; intervention not indicated | Moderate; persistent; psychosocial sequelae | - | - | - |
| Definition: A disorder characte | rized by a state of excessive gas in | the alimentary canal. | | <b>I</b> | |
| Gastric fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | n between the stomach and anoth | er organ or anatomic site. | T | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the gastric wa | all. | <u> </u> | | |
| Gastric necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | • | I . | 1 | 1 | |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation Definition: A disorder character | -<br>rized by a rupture in the stomach wa | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | 1 | | Soverely altered Cl function: | Life threatening consequences: | Death |
| Gastric stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Deam |
| Definition: A disorder character | rized by a narrowing of the lumen of | the stomach. | _ | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a circumscribed, inflammato | ry and necrotic erosive lesion on | the mucosal surface of the stomac | | |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by inflammation of the stomach | l. | T | T | |
| Gastroesophageal reflux<br>disease | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | rized by reflux of the gastric and/or d<br>y result in injury to the esophageal m | | | nd usually caused by incompetend | e of the lov |
| Gastrointestinal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site. | |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the gastrointestinal region | ٦. | | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to<br>maintain nutrition with dietary<br>and lifestyle modifications; may<br>need pharmacologic<br>intervention | Weight loss; refractory to medical intervention; unable to maintain nutrition orally | | - |
| Definition: A disorder character | rized by an incomplete paralysis of th | ne muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small inte | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to aliment orally | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the gingival region. | T | T | |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the hemorrho | ids. | T | T | |
| Hemorrhoids | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder character | rized by the presence of dilated veins | s in the rectum and surrounding a | rea. | | |
| leal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between the ileum and another o | organ or anatomic site. | | |
| lleal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | t e | 1 | 1 - 1 | 1 | |

| Gastrointestinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| | | | | | Ι. |
| Adverse Event | 1 | 2 | 3 | 4 | |
| leal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents in the ile | eum. | | |
| lleal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a rupture in the ileal wall. | _ | | | |
| lleal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by a narrowing of the lumen of | the ileum. | Т | T | |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the ileum. | | |
| lleus<br>Definition: A disorder characteri: | -<br>zed by failure of the ileum to transp | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Intra-abdominal hemorrhage | - | Medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by bleeding in the abdominal c | avity. | 1. | ı | ' |
| Jejunal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ।<br>zed by an abnormal communicatio। | ।<br>n between the ieiunum and anoth | 1 | I | 1 |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ਾ<br>zed by bleeding from the jejunal wa | all. | 1 ' | ı | 1 |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents in the je | ejunum. | | |
| Jejunal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ਾ<br>zed by a rupture in the jejunal wall. | · | · | ·<br> | |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a narrowing of the lumen of | the jejunum. | | | |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the jejunun | n. | · |
| Lip pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Lower gastrointestinal | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| hemorrhage | | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | l | cauterization indicated | operative intervention indicated | | ļ |
| Definition: A disorder characte | erized by bleeding from the lower gas | strointestinal tract (small intestine, | large intestine, and anus). | Т | 1 |
| Malabsorption | - | Altered diet; oral intervention indicated | Inability to aliment adequately;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inadequate absorption of nu | trients in the small intestine. Sym | ptoms include abdominal marked | discomfort, bloating and diarrhea. | |
| Mucositis oral | Asymptomatic or mild | Moderate pain; not interfering | Severe pain; interfering with oral | Life-threatening consequences; | Death |
| | symptoms; intervention not | with oral intake; modified diet | intake | urgent intervention indicated | |
| | indicated | indicated | | | |
| Definition: A disorder characte | erized by inflammation of the oral mu | cosal. | | 1 | |
| Nausea | Loss of appetite without | Oral intake decreased without | Inadequate oral caloric or fluid | - | - |
| | alteration in eating habits | significant weight loss, | intake; tube feeding, TPN, or | | |
| | | dehydration or malnutrition | hospitalization indicated | | |
| | erized by a queasy sensation and/or | | | | |
| estruction gastric | Asymptomatic; clinical or | Symptomatic; altered GI | Hospitalization indicated; | Life-threatening consequences; | Death |
| | diagnostic observations only; | function; limiting instrumental | elective operative intervention | urgent operative intervention | |
| | intervention not indicated ADL indicated; limiting self care ADL; disabling indicated | | | | |
| Definition: A disorder characte | ।<br>erized by blockage of the normal flow | of the contents in the stomach | 1 | I | I. |
| | | | Soverely altered Cl function | Life threatening sensesure | Dooth |
| Oral cavity fistula | Asymptomatic; clinical or diagnostic observations only; | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated; | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | intervention not indicated | Turiction | elective operative intervention | digent intervention indicated | |
| | | | indicated | | |
| Definition: A disorder characte | erized by an abnormal communication | n between the oral cavity and ano | ther organ or anatomic site. | ! | • |
| Oral dysesthesia | Mild discomfort; not interfering | Moderate pain; interfering with | Disabling pain; tube feeding or | _ | _ |
| oran ayoooanoona | with oral intake | oral intake | TPN indicated | | |
| Definition: A disorder characte | erized by a burning or tingling sensati | on on the lips, tongue or entire m | outh. | ı | 1 |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| oral nome.mage | ma, merremen net maleate a | intervention or minor | endoscopic, or elective | urgent intervention indicated | D Guill |
| | | cauterization indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by bleeding from the mouth. | • | • | | • |
| Oral pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | · . | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the mouth, tongue or lips | ' | ! | |
| Pancreatic duct stenosis | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| | diagnostic observations only; | function | tube feeding or hospitalization | urgent operative intervention | |
| | intervention not indicated | | indicated; elective operative | indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the pancreatic duct. | | | |
| Pancreatic fistula | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| | diagnostic observations only; | function | tube feeding or TPN or | urgent operative intervention | |
| | intervention not indicated | | hospitalization indicated; | indicated | |
| | | | elective operative intervention | | |
| | | | indicated | | 1 |
| Definition: A disorder characte | erized by an abnormal communication | n between the pancreas and anot | her organ or anatomic site. | 1 | , |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| | | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | | cauterization indicated | operative intervention indicated | l | l |
| Definition: A disorder characte | erized by bleeding from the pancreas | T | | Т | _ |
| Pancreatic necrosis | - | - | Tube feeding or TPN indicated; | Life-threatening consequences; | Death |
| | | | radiologic, endoscopic, or | urgent operative intervention | |
| | | | operative intervention indicated | indicated | |
| Definition: A disorder characte | erized by a necrotic process occurring | g in the pancreas. | | | |
| Pancreatitis | - | Enzyme elevation or radiologic | Severe pain; vomiting; medical | Life-threatening consequences; | Death |
| | 1 | l | 1 | 1 | 1 |
| | | findings only | intervention indicated (e.g., | urgent intervention indicated | |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | zed by inflammation of the pancrea | S. | 1 | | |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or gingivitis; multiple sites of bleeding on probing; moderate bone loss | Spontaneous bleeding; severe bone loss with or without tooth loss; osteonecrosis of maxilla or mandible | - | - |
| Definition: A disorder in the ging | ival tissue around the teeth. | 1 | | | |
| Peritoneal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a necrotic process occurring | in the peritoneum. | 1 | | |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by inflammation of the rectum. | | | | |
| Rectal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | n between the rectum and another | r organ or anatomic site. | | |
| Rectal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the rectal wal | and discharged from the anus. | | | |
| Rectal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by inflammation of the mucous | membrane of the rectum. | 1 | | |
| Rectal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents in the re | ctum. | | |
| Rectal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by a sensation of marked disco | omfort in the rectal region. | 1 | | |
| Rectal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by a rupture in the rectal wall. | T | 1 | | ı |
| Rectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a narrowing of the lumen of | the rectum. | T. | | |
| Rectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function (e.g. altered dietary<br>habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Retroperitoneal hemorrhage | -<br>ted by bleeding from the retroperite | Self-limited; intervention indicated | Transfusion, medical, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | | | Aguta galiyany gland negrasis: | Life threatening concequences: | Death |
| Salivary duct inflammation | Slightly thickened saliva; slightly altered taste (e.g., metallic) | markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis;<br>severe secretion-induced<br>symptoms (e.g., thick saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated;<br>limiting self care ADL; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the salivary | duct. | | | |
| Salivary gland fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe pain; interfering with oral<br>intake; tube feeding, TPN or<br>hospitalization indicated; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the intestinal contents. | _ | | |
| Small intestinal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the small intesti | ne wall. | | | |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the small intestine. | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on t | the mucosal surface of the small in | testine. | |
| Stomach pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the stomach. | 1 | | 1 |
| Γooth development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with oral surgery | Maldevelopment with impairment not surgically correctable; disabling | - | - |
| Definition: A disorder characteriz | red by a pathological process of the | e teeth occurring during tooth deve | elopment. | | |
| Γooth discoloration | Surface stains | - | - | - | - |
| Definition: A disorder characteriz | ted by a change in tooth hue or tint | t.<br>T | 1 | | |
| Toothache | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | l - | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Typhlitis | - | - | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal signs | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the cecum. | | | | |
| Upper gastrointestinal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the upper gas | trointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | |
| Vomiting | 1 - 2 episodes (separated by 5 minutes) in 24 hrs | 3 - 5 episodes (separated by 5 minutes) in 24 hrs | >=6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the reflexive act of ejecting t | he contents of the stomach throug | gh the mouth. | • | |
| Gastrointestinal disorders -<br>Other, specify | , , , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | disorders and administra | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold; | Moderate tremor of the entire | Severe or prolonged, not | - | - |
| Definition: A disorder charac | shivering; chattering of teeth<br>cterized by a sensation of cold that ofte | body; narcotics indicated<br>n marks a physiologic response to | responsive to narcotics sweating after a fever. | I | ļ |
| Death neonatal | - | = | - | = | Death |
| Definition: A disorder charac | cterized by cessation of life occurring d | uring the first 28 days of life. | I | | <u>'</u> |
| Death NOS | - | - | - | - | Death |
| Definition: A cessation of life | e that cannot be attributed to a CTCAE | term associated with Grade 5. | | | |
| Edema face | Localized facial edema | Moderate localized facial edema; limiting instrumental ADL | Severe swelling; limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by swelling due to excessive flo | uid accumulation in facial tissues. | 1 | 1 | |
| Edema limbs | 5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection | >10 - 30% inter-limb<br>discrepancy in volume or<br>circumference at point of<br>greatest visible difference;<br>readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | >30% inter-limb discrepancy in<br>volume; gross deviation from<br>normal anatomic contour;<br>limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by swelling due to excessive flu | uid accumulation in the upper or lo | wer extremities. | | |
| Edema trunk | Swelling or obscuration of anatomic architecture on close inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | Gross deviation from normal<br>anatomic contour; limiting self<br>care ADL | - | - |
| Facial pain | cterized by swelling due to excessive fli<br>Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Definition: A disorder charac | ।<br>cterized by a sensation of marked disco | 1 | J. 102 | l | 1 |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest;<br>limiting instrumental ADL | Fatigue not relieved by rest, limiting self care ADL | - | - |
| Definition: A disorder charac | cterized by a state of generalized weak | ness with a pronounced inability to | summon sufficient energy to acc | omplish daily activities. | |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>104.0 degrees F) for <=24 hrs | >40.0 degrees C (>104.0 degrees F) for >24 hrs | Death |
| Definition: A disorder charac | cterized by elevation of the body's temp | perature above the upper limit of n | ormal. | | |
| Flu like symptoms | Mild flu-like symptoms present | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder character cough. | cterized by a group of symptoms simila | r to those observed in patients wit | n the flu. It includes fever, chills, b | ody aches, malaise, loss of appet | ite and dry |
| Gait disturbance | Mild change in gait (e.g., wide-based, limping or hobbling) | Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL | Disabling; limiting self care ADL | - | - |
| | cterized by walking difficulties. | | | | T |
| Hypothermia | - | 35 - >32 degrees C; 95 - >89.6 degrees F | 32 - >28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C; 82.4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>hypotension, pulmonary edema,<br>acidemia, ventricular fibrillation) | |

| | Jonetan | disorders and administra | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Infusion related reaction | Mild transient reaction; infusion | Therapy or infusion interruption | Prolonged (e.g., not rapidly | Life-threatening consequences; | Death |
| illiusion relateu reaction | interruption not indicated; | indicated but responds promptly | responsive to symptomatic | urgent intervention indicated | Death |
| | intervention not indicated | to symptomatic treatment (e.g., | medication and/or brief | argone intervention indicated | |
| | miler verifier riet maleated | antihistamines, NSAIDS, | interruption of infusion); | | |
| | | narcotics, IV fluids); prophylactic | | | |
| | | medications indicated for <=24 | following initial improvement; | | |
| | | hrs | hospitalization indicated for | | |
| | | | clinical sequelae | | |
| Definition: A disorder characteriz | ।<br>zed by adverse reaction to the infus | ।<br>sion of pharmacological or biologic | | I | 1 |
| Infusion site extravasation | , | Erythema with associated | Ulceration or necrosis; severe | Life-threatening consequences; | Death |
| asien site sati a rasation | | symptoms (e.g., edema, pain, | tissue damage; operative | urgent intervention indicated | Dou |
| | | induration, phlebitis) | intervention indicated | angent intervention indicated | |
| Definition: A disorder characteria | ।<br>zed by leakage of a pharmacologic | | ' | I<br>selle. Signs and symptoms include | l<br>e induratio |
| | sation and marked discomfort at the | • | illusion site into the surrounding the | ssue. Olgris and symptoms include | e induranc |
| Injection site reaction | Tenderness with or without | Pain; lipodystrophy; edema; | Ulceration or necrosis; severe | Life-threatening consequences; | Death |
| • | associated symptoms (e.g., | phlebitis | tissue damage; operative | urgent intervention indicated | |
| | warmth, erythema, itching) | · | intervention indicated | | |
| Definition: A disorder characteriz | zed by an intense adverse reaction | (usually immunologic) developing | ' | I | 1 |
| Irritability | Mild; easily consolable | Moderate; limiting instrumental | Severe abnormal or excessive | _ | _ |
| Пітаріііту | ivilia, casily corisolable | ADL; increased attention | response; limiting self care ADL; | | - |
| | | indicated | inconsolable | | |
| 5 5 W A II A II A I | | ļ | 1 | l | 1 |
| Definition: A disorder characterize | zed by an abnormal responsivenes | s to stimuli or physiological arousa | ar; may be in response to pain, ing | nt, a drug, an emotional situation o | or a medic |
| Localized edema | Localized to dependent areas, | Moderate localized edema and | Severe localized edema and | - | _ |
| | no disability or functional | intervention indicated; limiting | intervention indicated; limiting | | |
| | impairment | instrumental ADL | self care ADL | | |
| Definition: A disorder characterize | red by swelling due to excessive flu | ı | 1 | I | 1 |
| Malaise | Uneasiness or lack of well being | | _ | | _ |
| Walaioo | Onedomes of lack of won being | being; limiting instrumental ADL | | | |
| Definition: A disorder characteriz | ed by a feeling of general discomf | | ı<br>feelina. | l | 1 |
| Multi-organ failure | | _ | Shock with azotemia and acid- | Life-threatening consequences | Death |
| Wali Organ landro | | | base disturbances; significant | (e.g., vasopressor dependent | Bouiii |
| | | | coagulation abnormalities | and oliguric or anuric or | |
| | | | coagulation abnormalities | ischemic colitis or lactic | |
| | | | | acidosis) | |
| Definition: A disorder characteriz | ed by progressive deterioration of | l<br>the lungs liver kidney and clotting | l<br>n mechanisms | / | 1 |
| Neck edema | Asymptomatic localized neck | Moderate neck edema; slight | Generalized neck edema (e.g., | _ | I . |
| veck edema | edema | obliteration of anatomic | difficulty in turning neck); | | - |
| | odoma | | limiting self care ADL | | |
| | | Handmarks: limiting instrumental | | | |
| | | landmarks; limiting instrumental ADL | Infiniting Sch care ADE | | |
| Definition: A disorder characteriz | ted by swelling due to an accumula | ADL | | | |
| | | ADL ation of excessive fluid in the neck | | - | <br> - |
| | ted by swelling due to an accumula | ADL | | - | - |
| Non-cardiac chest pain | | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Non-cardiac chest pain<br>Definition: A disorder characteriz | Mild pain | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Non-cardiac chest pain<br>Definition: A disorder characteriz | Mild pain | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. | Severe pain; limiting self care | - | - |
| Non-cardiac chest pain<br>Definition: A disorder characteriz<br>Pain | Mild pain | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL Severe pain; limiting self care | - | - |
| Non-cardiac chest pain<br>Definition: A disorder characteriz<br>Pain<br>Definition: A disorder characteriz | Mild pain<br>ted by discomfort in the chest unrel<br>Mild pain | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL Severe pain; limiting self care | - | - Death |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS | Mild pain<br>ted by discomfort in the chest unrel<br>Mild pain | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. | Severe pain; limiting self care ADL Severe pain; limiting self care ADL | - | - Death |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS Definition: An unexpected cessa | Mild pain ted by discomfort in the chest unrel Mild pain ted by the sensation of marked disc | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. | Severe pain; limiting self care ADL Severe pain; limiting self care ADL | - Life-threatening consequences; | - Death |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS Definition: An unexpected cessa General disorders and | Mild pain red by discomfort in the chest unred Mild pain red by the sensation of marked disc - tion of life that cannot be attributed | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. | · | '<br> |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS Definition: An unexpected cessa General disorders and administration site conditions - | Mild pain red by discomfort in the chest unred Mild pain red by the sensation of marked disc - tion of life that cannot be attributed Asymptomatic or mild | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL ated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. to a CTCAE term associated with | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant | Life-threatening consequences; | '<br> |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS | Mild pain red by discomfort in the chest unrel Mild pain red by the sensation of marked disc - tion of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately life- | Life-threatening consequences; | · |
| Non-cardiac chest pain Definition: A disorder characteriz Pain Definition: A disorder characteriz Sudden death NOS Definition: An unexpected cessa General disorders and administration site conditions - | Mild pain red by discomfort in the chest unrel Mild pain red by the sensation of marked disc - tion of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention indicated; limiting age- | Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately life-threatening; hospitalization or | Life-threatening consequences; | '<br> |

| Hepatobiliary disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bile duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Severely altered GI function;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a narrowing of the lumen of | the bile duct. | | | |
| Biliary fistula | - | Symptomatic and intervention not indicated | Severely altered GI function;<br>TPN indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by an abnormal communication | n between the bile ducts and anoth | ner organ or anatomic site. | T | |
| Cholecystitis | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by inflammation involving the g | allbladder. It may be associated w | vith the presence of gallstones. | | |
| Gallbladder fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Symptomatic or severely altered<br>GI function; TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | between the gallbladder and and | ther organ or anatomic site. | | |
| Gallbladder necrosis | - | - | - | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characterization | zed by a necrotic process occurring | g in the gallbladder. | T | T | |
| Gallbladder obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | zed by blockage of the normal flow | | | | |
| Gallbladder pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | omfort in the gallbladder region. | ' | ' | • |
| Gallbladder perforation | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a rupture in the gallbladder | wall. | | | I <sub>D</sub> ,, |
| Hepatic failure | - | - | Asterixis; mild encephalopathy; limiting self care ADL | Moderate to severe encephalopathy; coma; life-threatening consequences | Death |
| | zed by the inability of the liver to me | etabolize chemicals in the body. L | aboratory test results reveal abnor | rmal plasma levels of ammonia, bi | lirubin, lact |
| dehydrogenase, and alkaline ph | 1 | 0 , " " : | _ , | ler a | <b>.</b> |
| Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the liver. | | | | |
| Hepatic necrosis | - | - | - | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder characteriz | zed by a necrotic process occurring | g in the hepatic parenchyma. | | | |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | omfort in the liver region. | <b>.</b> | <b>.</b> | |
| Perforation bile duct | - | - | Radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Portal hypertension | - | Decreased portal vein flow | Reversal/retrograde portal vein flow; associated with varices and/or ascites | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an increase in blood pressu | re in the portal venous system. | | | |
| Portal vein thrombosis | - | Intervention not indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by the formation of a thrombus | (blood clot) in the portal vein. | | | |
| Hepatobiliary disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| | | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug fever <38 degrees C (<100.4 degrees F); intervention not indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an adverse local or general | response from exposure to an alle | | | I |
| Anaphylaxis | - | - | Symptomatic bronchospasm, with or without urticaria; parenteral intervention indicated; allergy-related edema/angioedema; hypotension | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an acute inflammatory react<br>resents with breathing difficulty, di | • | | | ypersensitivi |
| | | | | | Dooth |
| Autoimmune disorder | Asymptomatic; serologic or<br>other evidence of autoimmune<br>reaction, with normal organ<br>function; intervention not<br>indicated | Evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder resulting fr tissue constituents. | om loss of function or tissue destru | ction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individe | ual to his ow |
| Cytokine release syndrome | Mild reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | following initial improvement;<br>hospitalization indicated for<br>clinical sequelae (e.g., renal<br>impairment, pulmonary<br>infiltrates) | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| Definition: A disorder characterize | red by nausea, headache, tachyca | rdia, hypotension, rash, and shorti | ness of breath; it is caused by the | release of cytokines from the cells | i. |
| Serum sickness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash, urticaria, antihistamines indicated | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV<br>fluids indicated | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| | red by a delayed-type hypersensiti<br>e foreign antigen. Symptoms inclu | | | | |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | ving the abdominal cavity. | | 1 | |
| Anorectal infection | Localized; local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invo | ving the anal area and the rectum. | IV antibiotic antifungal or | Life threatening consequences: | Death |
| Appendicitis | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Deam |
| | rized by acute inflammation to the | | 1 | | Б. " |
| Appendicitis perforated | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by acute inflammation to the<br>iceal wall rupture causes the releas | vermiform appendix caused by a pa | athogenic agent with gangrenous o | changes resulting in the rupture of | the |
| Arteritis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | ving an artery. | | ·<br> | |
| Biliary tract infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the biliary tract. | 1 | ı | |
| Bladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invo | ving the bladder. | | | |
| Bone infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invo | | <u> </u> | I | L |
| Breast infection | - | Local infection with moderate<br>symptoms; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | Severe infection; axillary<br>adenitis; IV antibacterial,<br>antifungal, or antiviral<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | 1 | | I | L |
| Bronchial infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bronchi. | 1 | 1 | 1 |
| Catheter related infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process that | arises secondary to catheter use. | | | |
| Cecal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the cecum. | | | |
| Cervicitis infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| ا<br>Definition: A disorder characterize | ed by an infectious process involvi | ing the uterine cervix. | | ' | , |
| Conjunctivitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the conjunctiva. Clinical manife | estations include pink or red color | in the eyes. | 1 |
| Corneal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the cornea. | • | | |
| Cranial nerve infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing a cranial nerve. | | • | |
| Device related infection | - | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the use of a medical device. | T | T | |
| Duodenal infection | - | Moderate symptoms; medical intervention indicated (e.g., oral antibiotics) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the duodenum. | | | |
| Encephalitis infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>severe changes in mental<br>status; self-limited seizure<br>activity; focal neurologic<br>abnormalities | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the brain tissue. | | | |
| Encephalomyelitis infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the brain and spinal cord tissu | es. | · | ·<br> |
| Endocarditis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the endocardial layer of the he | art. | T | |
| John Maria Francisco | | | | | |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Enterocolitis infectious | - | Passage of >3 unformed stools<br>per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal<br>pain | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated;<br>profuse watery diarrhea with<br>signs of hypovolemia; bloody | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ted by an infectious process involv | ing the small and large intestines | diarrhea; fever; severe<br>abdominal pain; hospitalization<br>indicated | | |
| | Sa by an inconsas process involv | Local intervention indicated | IV antibiotic, antifungal, or | Life threatening concequences: | Death |
| Esophageal infection | - | (e.g., oral antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the esophagus. | | | |
| Eye infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated;<br>enucleation | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the eye. | | | |
| Gallbladder infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the gallbladder. | · | | |
| Gum infection | Local therapy indicated (swish and swallow) | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the gums. | | | |
| Hepatic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the liver. | | | |
| Hepatitis viral | Asymptomatic, treatment not indicated | - | Symptomatic liver dysfunction;<br>fibrosis by biopsy; compensated<br>cirrhosis; reactivation of chronic<br>hepatitis | Decompensated liver function<br>(e.g., ascites, coagulopathy,<br>encephalopathy, coma) | Death |
| Definition: A disorder characteriz | ed by a viral pathologic process in | volving the liver parenchyma. | T | <u> </u> | |
| Infective myositis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the skeletal muscles. | | | |
| Joint infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); needle aspiration indicated (single or multiple) | Arthroscopic intervention indicated (e.g., drainage) or arthrotomy (e.g., open surgical drainage) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | 1 | • | • | • |
| Kidney infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | T . | I . | 1 -r - auto manated | l | I . |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | T | Grade | T | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| .aryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an inflammatory process in | volving the larynx. | 1 | | |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characte | rized by an infectious process invol | ving the lips. | • | | |
| Lung infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | ving the lungs. | T | 1 | |
| Lymph gland infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | ving the lymph nodes. | I | I | |
| Mediastinal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the mediastinum. | I | 1 | _ |
| Meningitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by acute inflammation of the r | neninges of the brain and/or spinal | cord. | ' | • |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving a mucosal surface. | | | |
| Nail infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| | rized by an infectious process invol | | | | |
| Otitis externa | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process involuptoms include fullness, itching, swe | • | • | ive water exposure (swimmer's ea | r infection |
| Otitis media | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the middle ear. | | | |
| Ovarian infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | I | 1 | Intervention indicated | I | 1 |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involv | ing the pancreas. | | | |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | erized by an eruption consisting of pa | | | | o, and upper |
| | this rash does not present with whiteh | | İ | esions. | |
| Paronychia | Nail fold edema or erythema;<br>disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical intervention or IV antibiotics indicated; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by an infectious process involvi | ing the soft tissues around the nai | l. | _ | |
| Pelvic infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by an infectious process involving | ing the pelvic cavity. | T | T | 1 |
| Penile infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involvi | ing the penis. | | | |
| Periorbital infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by an infectious process involvi | | D/ | if_ | D#h |
| Peripheral nerve infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by an infectious process involvi | ing the peripheral nerves. | | Ī | |
| Peritoneal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by an infectious process involvi | ing the peritoneum. | 1 | 1 | 1 |
| Pharyngitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the throat. | | | | |
| Phlebitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| 1 | | Grade | | |
|---|---|---|---|---|
| | _ | | | |
| d bu an infactious process involuin | 2 | 3 | 4 | 5 |
| by an injectious process involving | ng the vein. Clinical manifestation | s include erythema, marked disco | mfort, swelling, and induration alo | ng the course |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| , | • . | N/ (2) (2) | | D " |
| | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| d by an infectious process involving | ng the prostate gland. | | | |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| d by a circumscribed and elevated | d skin lesion filled with pus. | | | |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | - | - | - |
| d by an infectious process involvir | ng the nasal mucosal. | | | |
| | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| d by an infectious process involvir | ng the salivary gland. | | • | |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| d by an infectious process involvir | ng the scrotum. | | | |
| - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| d by the presence of pathogenic r | nicroorganisms in the blood strea | m that cause a rapidly progressing | g systemic reaction that may lead | to shock. |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| d by an infectious process involving | ng the mucous membranes of the | paranasal sinuses. | | |
| | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| d by an infectious process involving | ng the skin. | Ī | Ī | |
| | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| d by an infectious process involving | ng the small intestine. | | | |
| | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| n by an intectious process involvir | ng soft tissues. | | | |
| - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | by an infectious process involving calized, local intervention indicated. | indicated (e.g., topical antibiotic, antifungal, or antiviral) by an infectious process involving the pleura. | Indicated (e.g., topical antibiotic, antifurgal, or antiviral) Iby an infectious process involving the pleura. Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) Iby an infectious process involving the prostate gland. Localized; local intervention indicated (e.g., antibiotic, antifungal, or antiviral) Iby an infectious process involving the prostate gland. Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Iby a circumscribed and elevated skin lesion filled with pus. Localized; local intervention indicated (e.g., antibiotic, antifungal, or antiviral) Iby an infectious process involving the nasal mucosal. Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, or antiviral) Iby an infectious process involving the salivary gland. Localized; local intervention indicated (e.g., antibiotic, antifungal, or antiviral) Localized; local intervention indicated (e.g., antibiotic, antifungal, or antiviral intervention indicated; radiologic or operative intervention indicated (e.g., antibiotic, antifungal, or antiviral intervention indicated (e.g., antibiotic, antifungal, or antiviral intervention indicated (e.g., antibiotic, antifungal, or antiviral intervention indicated (e.g., antibiotic, antifungal, or antiviral intervention indicated (e.g., antibiotic, antifungal, or antiviral intervention indicated (e.g., antibiotic, antifungal, or antiviral) Localized; local intervention indicated (e.g., antibioti | indicated (e.g., topical antibiotic, antifungal, or antiviral) antiviral intervention indicated (by an infectious process involving the pleura. Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) antibiotic, antifungal, antiviral intervention indicated (e.g., antibiotic, antifungal, antiviral) antiviral intervention indicated (e.g., topical antibiotic, antifungal, or antiviral intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) antiviral intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) intervention indicated (e.g., topical antibiotic, anti |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | Localized, local intervention indicated | oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing a stoma (surgically created op | ening on the surface of the body). | | |
| Tooth infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing a tooth. | I | 1 | |
| Tracheitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | 1 | Τ | T | |
| Upper respiratory infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the upper respiratory tract (nos | se, paranasal sinuses, pharynx, la | rynx, or trachea). | |
| Urethral infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the urethra. | | | |
| Urinary tract infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the urinary tract, most commo | nly the bladder and the urethra. | | |
| Uterine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the endometrium. It may exten | Id to the myometrium and parame | trial tissues. | • |
| Vaginal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the vagina. | | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the vulva. | | | |
| Wound infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the wound. | | | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | , | , poisoning and procedu | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention | Limiting instrumental ADL; | Limiting self care ADL; elective | | _ |
| | indicated | operative intervention indicated | surgery indicated | | |
| Definition: A finding of damage affected leg and foot. | to the ankle joint characterized by a | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | y moving th |
| Aortic injury | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | | | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage | to the aorta. | | I | indicated | l |
| Arterial injury | Asymptomatic diagnostic | Symptomatic (e.g., | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| ,, | finding; intervention not indicated | claudication); repair or revision<br>not indicated | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage | to an artery. | 1 | I | | l |
| Biliary anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | • . | |
| | not indicated | | intervention indicated | indicated | |
| | of bile due to breakdown of a biliary | | | • | |
| Bladder anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | of urine due to breakdown of a blad | lder anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | 1 |
| Bruising | Localized or in a dependent area | Generalized | - | - | - |
| Definition: A finding of injury of | the soft tissues or bone characteriz | ed by leakage of blood into surrou | nding tissues. | | 1 |
| Burn | Minimal symptoms; intervention not indicated | Medical intervention; minimal debridement indicated | Moderate to major debridement or reconstruction indicated | Life-threatening consequences | Death |
| • . | integrity to the anatomic site of an edepends on the length and intensi | | • • | nicals, direct heat, electricity, flame | es and |
| Dermatitis radiation | Faint erythema or dry | Moderate to brisk erythema; | Moist desquamation in areas | Life-threatening consequences; | Death |
| Joinnattia radiation | desquamation | patchy moist desquamation, | other than skin folds and | skin necrosis or ulceration of full | Death |
| | | mostly confined to skin folds | creases; bleeding induced by | thickness dermis; spontaneous | |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin graft indicated | |
| Definition: A finding of cutaneou | ।<br>is inflammatory reaction occurring a | I<br>as a result of exposure to biologica | I<br>ally effective levels of ionizing radia | 10 | l |
| Esophageal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| . 0 | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | |
| Definition: A finding of leakage | due to breakdown of an esophagea | al anastomosis (surgical connection | of two separate anatomic structu | res). | |
| Fall | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding of sudden r | novement downward, usually result | ting in injury. | T | | 1 |
| Fallopian tube anastomotic leak | diagnostic observations only; | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative | Life-threatening consequences; urgent operative intervention | Death |
| Definition: A finding of lookage | intervention not indicated | a anastamasis (auraical connectio | intervention indicated | indicated | |
| Fallopian tube perforation | due to breakdown of a fallopian tub | Symptomatic and intervention | | | Dooth |
| -allopian tube perforation | Asymptomatic diagnostic observations only; intervention not indicated | not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture of | f the fallopian tube wall. | | | | |
| Fracture | Asymptomatic; clinical or | Symptomatic but non-displaced; | Severe symptoms; displaced or | Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated | immobilization indicated | open wound with bone exposure; disabling; operative | urgent intervention indicated | |

| | ,, | , poisoning and procedu | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic observations only; intervention | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative | Life-threatening consequences;<br>urgent operative intervention | Death |
| | not indicated | Intervention indicated | intervention indicated | indicated | |
| Deficialization of localization of | 1 | <br>+ | • | Indicated | l |
| | ue to breakdown of a gastric anas | | | | I |
| Gastrointestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| leak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage d | ue to breakdown of a gastrointesti | nal anastomosis (surgical connec | tion of two separate anatomic struc | ctures). | |
| Gastrointestinal stoma necrosis | - | Superficial necrosis; | Severe symptoms; | Life-threatening consequences; | Death |
| | | intervention not indicated | hospitalization or elective | urgent intervention indicated | |
| | | | operative intervention indicated | | |
| Definition: A finding of a necrotic | process occurring in the gastroint | estinal tract stoma. | • | | |
| | The second containing in the gapa on the | | C | Life the state of | |
| Hip fracture | - | Hairline fracture; mild pain; | Severe pain; hospitalization or | Life-threatening consequences; | - |
| | | limiting instrumental ADL; non-<br>surgical intervention indicated | intervention indicated for pain | symptoms associated with | |
| | | surgical intervention indicated | control (e.g., traction); operative intervention indicated | neurovascular compromise | |
| Distriction Associated to the control of the contro | I de la companya del companya de la companya del companya de la co | l | 1 | l | 1 |
| | injury to the hip in which the contir | nuity of either the femoral head, fe | emoral neck, intertrochanteric or su | 1 | 1 |
| Injury to carotid artery | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | | | care ADL (e.g., transient | urgent intervention indicated | |
| | | | cerebral ischemia); repair or | | |
| | | | revision indicated | | |
| Definition: A finding of damage to | the carotid artery. | | | | |
| Injury to inferior vena cava | - | - | - | Life-threatening consequences; | Death |
| | | | | urgent intervention indicated | |
| Definition: A finding of damage to | o the inferior vena cava | 1 | ' | | ' |
| | T T T T T T T T T T T T T T T T T T T | | Comptematic limiting celf care | Life threatening concessioness. | Dooth |
| Injury to jugular vein | - | <del>-</del> | Symptomatic limiting self care | Life-threatening consequences; | Death |
| | | | ADL; disabling; repair or | urgent intervention indicated | |
| | Į. | 1 | revision indicated | I | l |
| Definition: A finding of damage to | the jugular vein. | 1 | | 1 | |
| Injury to superior vena cava | Asymptomatic diagnostic | Symptomatic; repair or revision | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | finding; intervention not | not indicated | care ADL; disabling; repair or | evidence of end organ damage; | |
| | indicated | | revision indicated | urgent operative intervention | |
| | | | | indicated | |
| Definition: A finding of damage to | the superior vena cava. | | | | |
| Intestinal stoma leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage of | f contents from an intestinal stoma | s (surgically created opening on th | ue surface of the hody) | ' | ' |
| | . sssino irom ari intestinai stoma | ì | 1 | l ife threate-i | D" |
| Intestinal stoma obstruction | - | Self-limited; intervention not | Severe symptoms; IV fluids, | Life-threatening consequences; | Death |
| | | indicated | tube feeding, or TPN indicated | urgent operative intervention | |
| | | | >=24 hrs; elective operative | indicated | |
| | 1 | | intervention indicated | I | I |
| Definition: A finding of blockage | of the normal flow of the contents | of the intestinal stoma. | | T | 1 |
| Intestinal stoma site bleeding | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| | clinical exam; intervention not | intervention indicated | indicated; radiologic or | urgent intervention indicated | |
| | indicated | | endoscopic intervention | | |
| | | | indicated | | |
| Definition: A finding of blood leak | age from the intestinal stoma. | | | | |
| Intraoperative arterial injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| | organ/structure indicated | organ/structure indicated | reconstruction of injured | urgent intervention indicated | |
| | o.ganionaotaro maioatoa | S.ganion dotaro indicato | organ/structure indicated; | angent intervention indicated | |
| | | | disabling | | |
| Dofinition: A finding of down | on ortony during a series - L- | duro | <del></del> | I | ı |
| ווושם: A finding of damage to | o an artery during a surgical proce | | | | |
| | | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| Intraoperative breast injury | Primary repair of injured | - | | | |
| Intraoperative breast injury | organ/structure indicated | organ/structure indicated | reconstruction of injured | urgent intervention indicated | |
| Intraoperative breast injury | | - | | | |

| | J, | , poisoning and proced | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | the breast parenchyma during a | | • | • | |
| Intraoperative cardiac injury | - | - | Primary repair of injured organ/structure indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the heart during a surgical proce | edure. | | | |
| Intraoperative ear injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection of injured organ/structure indicated; disabling (e.g., impaired hearing; impaired balance) | Life-threatening consequences; urgent intervention indicated | Death |
| | o the ear during a surgical proced | | | | I |
| Intraoperative endocrine injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the endocrine gland during a sui | rgical procedure. | | | |
| Intraoperative gastrointestinal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the gastrointestinal system durin | g a surgical procedure. | | | |
| Intraoperative head and neck injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the head and neck during a surg | ical procedure. | | | |
| Intraoperative hemorrhage | - | - | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical proc | edure. | · | · | • |
| Intraoperative hepatobiliary injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the hepatic parenchyma and/or | biliary tract during a surgical pro | cedure. | | |
| Intraoperative musculoskeletal<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the musculoskeletal system duri | ng a surgical procedure. | | 1 | |
| Intraoperative neurological injury | Primary repair of injured organ/structure indicated the nervous system during a sur | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | | Ĭ | 0 11 " | 17.0 | Б. " |
| Intraoperative ocular injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the eye during a surgical proced | ure. | | 1 | |
| Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the kidney during a surgical prod | cedure. | | | |
| Intraoperative reproductive tract injury | | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of damage to | the reproductive organs during a | surgical procedure. | | | |
| ntraoperative respiratory injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the respiratory system during a s | urgical procedure. | | | |
| Intraoperative skin injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the skin during a surgical proced | ure. | | | |
| Intraoperative splenic injury | | Primary repair of injured organ/structure indicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the spleen during a surgical proc | | 0 | if_ 4 4i | D41- |
| Intraoperative urinary injury Definition: A finding of damage to | Primary repair of injured organ/structure indicated organ/structure indicated or the urinary system during a surg | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | | T . | Complete reception or | Life threatening concequences: | Death |
| Intraoperative venous injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Deam |
| Definition: A finding of damage to | a vein during a surgical procedu | e. | | | |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | urine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | indicated | Death |
| | | | f two separate anatomic structure | ĺ | L |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | indicated | Death |
| | | 1 | of two separate anatomic structure | 1 | 1_ |
| Postoperative hemorrhage Definition: A finding of bleeding of | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; radiologic, endoscopic, or operative intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Postoperative thoracic | ssang attor a surgiour procedur | Extubated within 24 - 72 hrs | Extubated >72 hrs | Life threatening circus | Death |
| Postoperative thoracic procedure complication | | postoperatively | postoperatively, but before tracheostomy indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A finding of a previous | ly undocumented problem that oc | curs after a thoracic procedure. | T | T | |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental<br>ADL | Severe symptoms; elective operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | I |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | of the intestinal stoma (surgically | | | | l |
| Prolapse of urostomy | Asymptomatic; clinical or | Local care or maintenance; | Dysfunctional stoma; elective | Life-threatening consequences; | Death |
| | diagnostic observations only; | minor revision indicated | operative intervention or major | urgent intervention indicated | |
| | intervention not indicated | | stomal revision indicated | | l |
| Definition: A finding of displacem | ent of the urostomy. | | T | <u> </u> | |
| Radiation recall reaction | Faint erythema or dry | Moderate to brisk erythema; | Moist desquamation in areas | Life-threatening consequences; | Death |
| (dermatologic) | desquamation | patchy moist desquamation, | other than skin folds and | skin necrosis or ulceration of full | |
| | | mostly confined to skin folds | creases; bleeding induced by | thickness dermis; spontaneous | |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin graft indicated | |
| Definition: A finding of courts okin | inflammatany reaction soused by | <br> | <br> | 1- | l<br>.to=room |
| - | inflammatory reaction caused by liting inflammatory reaction caused by liting inflammatory inflammatory inflammatory inflammatory. | | - | lowing radiotrierapy. The initamina | itory reac |
| · | 1 | | | | D41- |
| Rectal anastomotic leak | Asymptomatic diagnostic observations only; intervention | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative | Life-threatening consequences; urgent operative intervention | Death |
| | not indicated | intervention indicated | intervention indicated | indicated | |
| Definition: A finding of leakage de | ue to breakdown of a rectal anasto | I<br>amosis (surgical connection of two | ' | | I |
| <u> </u> | | | <u> </u> | | |
| Seroma | Asymptomatic; clinical or | Symptomatic; simple aspiration | Symptomatic, elective radiologic | - | - |
| | diagnostic observations only;<br>intervention not indicated | indicated | or operative intervention indicated | | |
| Definition A finding of towns 19 | 1 | I | majoatou | I | l |
| | collection of serum in the tissues. | | | I | |
| Small intestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| eak | observations only; intervention | intervention indicated | endoscopic or elective operative | | |
| | not indicated | l | intervention indicated | indicated | l |
| | ue to breakdown of an anastomosi | | arate anatomic structures) in the si | | |
| Spermatic cord anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| leak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage de | ue to breakdown of a spermatic co | ord anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Spinal fracture | Mild back pain; nonprescription | Moderate back pain; | Severe back pain; | Life-threatening consequences; | Death |
| | analgesics indicated | prescription analgesics | hospitalization or intervention | symptoms associated with | |
| | | indicated; limiting instrumental | indicated for pain control (e.g., | neurovascular compromise | |
| | | ADL | vertebroplasty); limiting self care ADL; disability | | |
| D-6-iti | | <br> | , , | ļ | l |
| | injury to the spine in which the con | | | | ı |
| Stenosis of gastrointestinal | - | Symptomatic; IV fluids indicated | Severely altered GI function; | Life-threatening consequences; | Death |
| stoma | | <24 hrs; manual dilation at<br>bedside | tube feeding, TPN or hospitalization indicated; | urgent operative intervention indicated | |
| | | bedside | elective operative intervention | indicated | |
| | | | indicated | | |
| Definition: A finding of parrowing | of the gastrointestinal stoma (surg | ı<br>rically created opening on the surf | ace of the body) | I . | 1 |
| Stomal ulcer | Asymptomatic; clinical or | Symptomatic; medical | Severe symptoms; elective | | |
| Storial dicei | diagnostic observations only; | intervention indicated | operative intervention indicated | - | - |
| | intervention not indicated | intervention indicated | operative intervention indicated | | |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ı<br>ırv and necrotic erosive lesion on t | ı<br>he jejunal mucosal surface close t | i<br>to the anastomosis site following a | 1 |
| gastroenterostomy procedure. | oa z, a onoamoonboa, milaminato | ., 110010110 0100110 1001011 011 1 | jojaniai maooodi sundoo olose l | .s and anadomodis site following a | |
| Tracheal hemorrhage | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| | clinical or diagnostic exam; | intervention indicated | indicated; radiologic or | urgent intervention indicated | |
| | intervention not indicated | | endoscopic intervention | | |
| | | | indicated | | |
| Definition: A finding of bleeding for | rom the trachea. | | | | |
| Fracheal obstruction | Partial asymptomatic | Symptomatic (e.g., noisy airway | Stridor; radiologic or endoscopic | Life-threatening airway | Death |
| | obstruction on examination | breathing), no respiratory | intervention indicated (e.g., | compromise; urgent intervention | Joann |
| | (e.g., visual, radiologic or | distress; medical intervention | stent, laser); limiting self care | indicated (e.g., tracheotomy or | |
| | endoscopic) | indicated (e.g., steroids); limiting | | intubation) | |
| | . , | instrumental ADL | | , | |
| | 1 | ļ | • | • | • |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Tracheostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood lea | kage from the tracheostomy site. | + | | | |
| Ureteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | lue to breakdown of a ureteral anas | T T | | T . | |
| Jrethral anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a urethral ana | stomosis (surgical connection of tw | vo separate anatomic structures). | | |
| Urostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | of contents from a urostomy. | | | Г | |
| Urostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or endoscopic repair or stent placement indicated | Altered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | <del>-</del> | | | |
| Urostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding | from the urostomy site. | ' | • | • | • |
| Urostomy stenosis | - | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | g of the opening of a urostomy. | | | | |
| Uterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a uterine anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a rupture in the uterine wall. | | | Lee al | ъ " |
| /aginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a vaginal anas | stomosis (surgical connection of tw | o separate anatomic structures). | 1 | |
| Vas deferens anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vas deferens | s anastomosis (surgical connection | n of two separate anatomic structu | res). | |
| Vascular access complication | - | Device dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including pulmonary embolism or life-threatening thrombus | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Venous injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated; disabling | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | a vein. | | | | |
| Wound complication | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound; local care indicated | Hernia without evidence of<br>strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by<br>operative intervention indicated | Hernia with evidence of<br>strangulation; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| Wound dehiscence | Incisional separation of <=25% | Incisional separation >25% of | Fascial disruption or dehiscence | Life-threatening consequences; | Death |
| wound deniscence | of wound, no deeper than superficial fascia | wound with local care;<br>asymptomatic hernia or<br>symptomatic hernia without<br>evidence of strangulation | without evisceration; primary wound closure or revision by operative intervention indicated | Lire-inreatening consequences;<br>symptomatic hernia with<br>evidence of strangulation;<br>fascial disruption with<br>evisceration; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| Definition: A finding of separation | of the approximated margins of a | surgical wound. | T | T | 1 |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of traumatic | injury to the wrist joint in which the | continuity of a wrist bone is broke | en. | | |
| Injury, poisoning and procedural complications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Investigations | <b>S</b> | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | y test result in which the partial th | | | possible indicator of coagulopat | hy, a prolonge |
| | may occur in a variety of disease | | | | |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | | 1 , | 1 | T |
| Alkaline phosphatase increased | 1 | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | | 1 | | |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen. | _ |
| Blood antidiuretic hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of antidiuretic horm | one in the blood specimen. | | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is as | ssociated with jaundice. | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotropl | hin in a blood specimen. | | • |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; | Symptomatic; medical intervention indicated; limiting | Severe symptoms; limiting self care ADL | - | - |
| | intervention not indicated | instrumental ADL | | | |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of gonadotrophin h | ormone in a blood specimen. | Т | 1 |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | l<br>bnormal levels of prolactin bormor | l<br>ne in a blood specimen | l | Ţ |
| Carbon monoxide diffusing | 1 | 6 - 8 units below LLN; for follow- | i i | _ | |
| capacity decreased | up, a decrease of 3 - 5 units (ml/min/mm Hg) below the baseline value | up, an asymptomatic decrease of >5 - 8 units (ml/min/mm Hg) below the baseline value | units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., >Grade 2 hypoxia or >Grade 2 or higher dyspnea) | | |
| Definition: A finding based on lun | g function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | | |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test resul | t which indicates increased levels | of cardiac troponin I in a biologica | l specimen. | T | |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with<br>myocardial infarction as defined<br>by the manufacturer | - | - |
| Definition: A laboratory test resul | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | | • |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 10e9="" 500="" <lln="" l<="" mm3;="" td="" x=""><td>&lt;500 - 200/mm3; &lt;0.5 - 0.2 x<br/>10e9 /L</td><td>&lt;200 - 50/mm3; &lt;0.2 x 0.05 -<br/>10e9 /L</td><td>&lt;50/mm3; &lt;0.05 x 10e9 /L</td><td>-</td></lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | · |
| Cholesterol high | | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | oratory test results that indicate h | igher than normal levels of cholest | terol in a blood specimen. | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in levels of creatine pho | osphokinase in a blood specimen | • | • |

| | | Investigations | <u> </u> | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of creatinine in a b | iological specimen. | <b>I</b> | |
| Ejection fraction decreased | - | Resting ejection fraction (EF) 50 - 40%; 10 - 19% drop from baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline | Resting ejection fraction (EF) <20% | - |
| Definition: The percentage compr<br>contraction. | uted when the amount of blood eje | ected during a ventricular contracti | on of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected interval prolonged | | QTc 481 - 500 ms | QTc >= 501 ms on at least two separate ECGs | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| | i i | bnormally long corrected QT inter | | | 1 |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75% decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of fibrinogen i | n a blood specimen. | ' | • |
| Forced expiratory volume decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on tes | t results that indicate a relative de | crease in the fraction of the forced | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate h | igher than normal levels of the enz | yme gamma-glutamyltransferase | in the blood specimen. GGT (gan | nma- |
| glutamyltransferase ) catalyzes th | ne transfer of a gamma glutamyl g | roup from a gamma glutamyl pept | ide to another peptide, amino acid | s or water. | |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of growth hormone | in a biological specimen. | | |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of haptoglobir | n in a blood specimen. | • | |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN | Increase in >4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | - | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of hemoglobin in a | biological specimen. | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation | >2.5 x ULN; >2.5 times above baseline if on anticoagulation | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the ratio of the patier | t's prothrombin time to a control s | ample in the blood. | |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of lipase in | a biological specimen. | | |
| Lymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of lymphocyte | es in a blood specimen. | | |
| Lymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormal increase in the numbe | r of lymphocytes in the blood, effu | sions or bone marrow. | |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of neutrophils | s in a blood specimen. | | |
| Pancreatic enzymes decreased | <lln and="" asymptomatic<="" td=""><td>Increase in stool frequency, bulk, or odor; steatorrhea</td><td>Sequelae of absorption deficiency</td><td>-</td><td>-</td></lln> | Increase in stool frequency, bulk, or odor; steatorrhea | Sequelae of absorption deficiency | - | - |
| D 6 11 | poratory test results that indicate a | n decrease in levels of nancreatic | ·<br>enzymes in a biological specimen. | | |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<="" 75,000="" <lln="" mm3;="" td=""><td>&lt;75,000 - 50,000/mm3; &lt;75.0 -</td><td>&lt;50,000 - 25,000/mm3; &lt;50.0 -</td><td>&lt;25,000/mm3; &lt;25.0 x 10e9 /L</td><td>-</td></lln> | <75,000 - 50,000/mm3; <75.0 - | <50,000 - 25,000/mm3; <50.0 - | <25,000/mm3; <25.0 x 10e9 /L | - |
| | 75.0 x 10e9 /L | 50.0 x 10e9 /L | 25.0 x 10e9 /L | | |
| Definition: A finding based on lab | poratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the levels of amylase | e in a serum specimen. | | |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | - |
| Definition: A finding based on tes | st results that indicate urine produc | ction is less relative to previous ou | tput. | | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value; | <50% of predicted value; | - | - |
| | | limiting instrumental ADL | limiting self care ADL | | |
| · | lmonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | num inhalation) when compared to | the predicted |
| value. | | T | T | | |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characterize | d by an increase in overall body w | eight; for pediatrics, greater than t | he baseline growth curve. | 1 | |
| Weight loss | 5 to <10% from baseline; | 10 - <20% from baseline; | >=20% from baseline; tube | - | - |
| | intervention not indicated | nutritional support indicated | feeding or TPN indicated | | |
| Definition: A finding characterize | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" td="" x<=""><td>&lt;3000 - 2000/mm3; &lt;3.0 - 2.0 x</td><td>&lt;2000 - 1000/mm3; &lt;2.0 - 1.0 x</td><td>&lt;1000/mm3; &lt;1.0 x 10e9 /L</td><td> -</td></lln> | <3000 - 2000/mm3; <3.0 - 2.0 x | <2000 - 1000/mm3; <2.0 - 1.0 x | <1000/mm3; <1.0 x 10e9 /L | - |
| | 10e9 /L | 10e9 /L | 10e9 /L | | |
| Definition: A finding based on lab | poratory test results that indicate a | n decrease in number of white blo | od cells in a blood specimen. | | |
| Investigations - Other, specify | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| cidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| efinition: A disorder characteriz | zed by abnormally high acidity (high | h hydrogen-ion concentration) of t | he blood and other body tissues. | T | |
| Alcohol intolerance | - | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterized in the comiting, indigestion and headage in the comiting in the community of the communi | zed by an increase in sensitivity to | the adverse effects of alcohol, wh | ich can include nasal congestion, | skin flushes, heart dysrhythmias, | nausea, |
| Alkalosis | pH >normal, but <=7.5 | | pH >7.5 | Life-threatening consequences | Death |
| | 1. | - | 1. | Life-tiffeaterining consequences | Death |
| | zed by abnormally high alkalinity (lo | | | Life 45 | D41- |
| Anorexia | Loss of appetite without alteration in eating habits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a loss of appetite. | | | | _ |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by excessive loss of water from | n the body. It is usually caused by | severe diarrhea, vomiting or diaph | noresis. | |
| Glucose intolerance | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an inability to properly metal | bolize glucose. | | | |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | zed by laboratory test results that ir | ,<br>ndicate an elevation in the concen | ration of calcium (corrected for all | oumin) in blood. | • |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz<br>ntolerance. | zed by laboratory test results that in | ndicate an elevation in the concen | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucose |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz<br>he use of diuretic drugs. | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of potassium in the blood; a | associated with kidney failure or so | ometimes w |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23<br>mmol/L | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that in | ndicate an elevation in the concen | tration of magnesium in the blood | T | |
| lypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterization | zed by laboratory test results that in | ndicate an elevation in the concen | tration of sodium in the blood. | Τ | T |
| lypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4 mmol/L;<br>life-threatening consequences | Death |
| efinition: A disorder characteriz | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of triglyceride concentration | n in the blood. | 1 |
| lyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| efinition: A disorder characteriz | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of uric acid. | | |
| lypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characterize | zed by laboratory test results that ir | ndicate a low concentration of albu | umin in the blood. | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -<br="">1.0 mmol/L</lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 - 6.0 mg/dL; <1.75 - 1.5 mmol/L; lonized calcium <0.9 - 0.8 mmol/L; hospitalization indicated | Corrected serum calcium of<br><6.0 mg/dL; <1.5 mmol/L;<br>Ionized calcium <0.8 mmol/L;<br>Iife-threatening consequences | Death |
| Definition: A disorder characterize | ed by laboratory test results that ir | ndicate a low concentration of calc | ium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0<br="" 55="" <lln="" dl;="" mg="">mmol/L</lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of gluc | ose in the blood. | | |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><pre><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" pre="" symptomatic;=""></lln></pre></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <pre><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" pre="" symptomatic;=""></lln></pre> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate a low concentration of pota | assium in the blood. | | |
| Hypomagnesemia | <lln -="" 0.5="" 1.2="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3 mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3 mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of mag | nesium in the blood. | | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate a low concentration of sod | um in the blood. | | |
| Hypophosphatemia | <lln -="" 0.8="" 2.5="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL; &lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 - 1.0 mg/dL; &lt;0.6 - 0.3<br/>mmol/L</td><td>&lt;1.0 mg/dL; &lt;0.3 mmol/L; life-<br/>threatening consequences</td><td>Death</td></lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6 mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3<br>mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of pho | sphates in the blood. | | |
| Iron overload | - | Moderate symptoms; intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by accumulation of iron in the ti | issues. | | | |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| Definition: A disorder characteriz | ed by having a high amount of boo | dy fat. | | | |
| Tumor lysis syndrome | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by metabolic abnormalities that | result from a spontaneous or the | rapy-related cytolysis of tumor cell | S | |
| Metabolism and nutrition disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the abdomir | nal wall. | | |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in a joint. | T | 1 | |
| Arthritis | Mild pain with inflammation, erythema, or joint swelling | Moderate pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inflammation involving a joir | it. | 1 | 1 | 1 |
| Avascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by necrotic changes in the bond<br>of the destruction of the bone struction | | d supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the back region. | | _ | |
| Bone pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the bones. | T | 1 | |
| Buttock pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the buttocks. | | | |
| Chest wall pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the chest wall region. | T | T | |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth o | of bone. | | | |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the | deep connective tissues. | 1 | 1 | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n on the lateral side of the body in | the region below the ribs and abo | ove the hip. | |
| Generalized muscle weakness | Symptomatic; weakness<br>perceived by patient but not<br>evident on physical exam | Symptomatic; weakness evident on physical exam; weakness limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | - |
| | ed by a reduction in the strength o | · . | | | Τ |
| Growth suppression | Reduction in growth velocity by 10 - 29% ideally measured over the period of a year ed by of stature that is smaller that | Reduction in growth velocity by 30 - 49% ideally measured over the period of a year or 0 - 49% reduction in growth from the baseline growth curve | Reduction in growth velocity of<br>>=50% ideally measured over<br>the period of a year | - | - |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Head soft tissue necrosis | - | Local wound care; medical | Operative debridement or other | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., | invasive intervention indicated | urgent intervention indicated | |
| | | dressings or topical | (e.g., tissue reconstruction, flap | | |
| | | medications) | or grafting) | | |
| Definition: A disorder characterize | ed by a necrotic process occurring | in the soft tissues of the head. | | ! | |
| Joint effusion | Asymptomatic; clinical or | Symptomatic; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL; elective operative | | |
| | intervention not indicated | in or arrivation at 7 to 2 | intervention indicated; disabling | | |
| Definition: ∆ disorder characteriz | ed by excessive fluid in a joint, usu | l<br>Ially as a result of joint inflammati | - 1 | l | l |
| | | >25 - 50% decrease in ROM; | >50% decrease in ROM; limiting | | |
| Joint range of motion decreased | | · · | , , | - | - |
| | motion); decreased ROM | limiting instrumental ADL | self care ADL; disabling | | |
| 5 5 W A P A A A A A A A A A A A A A A A A A | limiting athletic activity | · · · · · | | | l |
| | ed by a decrease in joint flexibility | | | | 1 |
| Joint range of motion decreased | Mild restriction of rotation or | Rotation <60 degrees to right or | Ankylosed/fused over multiple | - | - |
| cervical spine | flexion between 60 - 70 degrees | left; <60 degrees of flexion | segments with no C-spine | | |
| | 1 | | rotation | 1 | 1 |
| Definition: A disorder characterize | ed by a decrease in flexibility of a | cervical spine joint. | 1 | | |
| Joint range of motion decreased | Stiffness; difficulty bending to | Pain with range of motion | <50% lumbar spine flexion; | - | - |
| lumbar spine | the floor to pick up a very light | (ROM) in lumbar spine; requires | associated with symptoms of | | |
| | object but able to do athletic | a reaching aid to pick up a very | ankylosis or fused over multiple | | |
| | activity | light object from the floor | segments with no L-spine | | |
| | | | flexion (e.g., unable to reach to | | |
| | | | floor to pick up a very light | | |
| | | | object) | | |
| Definition: A disorder characterize | ·<br>ed by a decrease in flexibility of a l | lumbar spine joint. | , | ' | • |
| Kyphosis | Asymptomatic; clinical or | Moderate accentuation; limiting | Severe accentuation; operative | - | _ |
| ,, | diagnostic observations only; | instrumental ADL | intervention indicated; limiting | | |
| | intervention not indicated | | self care ADL | | |
| Definition: A disorder characterize | ed by an abnormal increase in the | curvature of the thoracic portion of | of the spine. | • | • |
| Lordosis | Asymptomatic; clinical or | Moderate accentuation; limiting | Severe accentuation; operative | - | - |
| | diagnostic observations only; | instrumental ADL | intervention indicated; limiting | | |
| | intervention not indicated | | self care ADL | | |
| Definition: A disorder characterize | ।<br>ed by an abnormal increase in the | curvature of the lumbar portion of | ' | l | 1 |
| Muscle weakness left-sided | Symptomatic; perceived by | Symptomatic; evident on | Limiting self care ADL; disabling | | |
| viuscie weakiless leit-sided | patient but not evident on | physical exam; limiting | Limiting sell care ADL, disabiling | - | - |
| | physical exam | instrumental ADL | | | |
| | 1 | l | l a badu | | l |
| D-fi-iti | | t the muscles on the left side of th | e boay. | | |
| Definition: A disorder characterize | | | | | |
| Definition: A disorder characterize Muscle weakness lower limb | Symptomatic; perceived by | Symptomatic; evident on | Limiting self care ADL; disabling | - | - |
| | Symptomatic; perceived by patient but not evident on | Symptomatic; evident on physical exam; limiting | | - | - |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | | - | - |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Muscle weakness lower limb Definition: A disorder characteriz | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on | | - | - |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting | Limiting self care ADL; disabling | - | - |
| Muscle weakness lower limb Definition: A disorder characterize | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on | Limiting self care ADL; disabling | - | - |
| Muscle weakness lower limb Definition: A disorder characterize Muscle weakness right-sided | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by patient but not evident on | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling Limiting self care ADL; disabling | - | - |
| Muscle weakness lower limb Definition: A disorder characteriz Muscle weakness right-sided Definition: A disorder characteriz | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling Limiting self care ADL; disabling | | - |
| Muscle weakness lower limb Definition: A disorder characterize Muscle weakness right-sided | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL f the muscles on the right side of the muscles on the right side of | Limiting self care ADL; disabling Limiting self care ADL; disabling he body. | | - |
| Muscle weakness lower limb Definition: A disorder characteriz Muscle weakness right-sided Definition: A disorder characteriz | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength o Symptomatic; perceived by | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL f the muscles on the right side of the Symptomatic; evident on | Limiting self care ADL; disabling Limiting self care ADL; disabling he body. | | - |
| Muscle weakness lower limb Definition: A disorder characterize Muscle weakness right-sided Definition: A disorder characterize Muscle weakness trunk | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL f the muscles on the right side of Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling Limiting self care ADL; disabling he body. | | - |
| Muscle weakness lower limb Definition: A disorder characterize Muscle weakness right-sided Definition: A disorder characterize Muscle weakness trunk Definition: A disorder characterize | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL f the muscles on the right side of the Symptomatic; evident on physical exam; limiting instrumental ADL f the trunk muscles. | Limiting self care ADL; disabling Limiting self care ADL; disabling the body. Limiting self care ADL; disabling | - | - |
| Muscle weakness lower limb Definition: A disorder characterize Muscle weakness right-sided Definition: A disorder characterize Muscle weakness trunk Definition: A disorder characterize | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by a reduction in the strength of Symptomatic; perceived by | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL f the muscles on the right side of the Symptomatic; evident on physical exam; limiting instrumental ADL f the trunk muscles. Symptomatic; evident on | Limiting self care ADL; disabling Limiting self care ADL; disabling he body. | - | - |
| Muscle weakness lower limb Definition: A disorder characterize Muscle weakness right-sided Definition: A disorder characterize Muscle weakness trunk | Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of Symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of symptomatic; perceived by patient but not evident on physical exam ed by a reduction in the strength of | Symptomatic; evident on physical exam; limiting instrumental ADL f the lower limb muscles. Symptomatic; evident on physical exam; limiting instrumental ADL f the muscles on the right side of the Symptomatic; evident on physical exam; limiting instrumental ADL f the trunk muscles. | Limiting self care ADL; disabling Limiting self care ADL; disabling the body. Limiting self care ADL; disabling | - | - |

| Musculoskeletal and connective tissue disorders Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or asymmetry able to be remediated by prosthesis (e.g., shoe insert) or covered by clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; disabling | - | - |
| Definition: A disorder character | ized by of a malformation of the mu | sculoskeletal system. | | | |
| Myalgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | , | |
| Myositis | Mild pain | Moderate pain associated with weakness; pain limiting instrumental ADL | Pain associated with severe weakness; limiting self care ADL | - | - |
| Definition: A disorder character | ized by inflammation involving the s | keletal muscles. | | | 1 |
| Neck pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | ized by marked discomfort sensatio | n in the neck area. Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | zed by a necrotic process occurring | in the soft tissues of the neck. | | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of osteoporosis or Bone Mineral Density (BMD) t-score -1 to -2.5 (osteopenia); no loss of height or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm;<br>hospitalization indicated; limiting<br>self care ADL | - | - |
| Definition: A disorder charactericomposition), resulting in increa | ized by reduced bone mass, with a ased fracture incidence. | decrease in cortical thickness and | I in the number and size of the trab | peculae of cancellous bone (but no | ormal cher |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensatio | n in the upper or lower extremities | S | | |
| Pelvic soft tissue necrosis | | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| | ized by a necrotic process occurring | , | | | |
| Scoliosis | <20 degrees; clinically undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | - | - |
| Definition: A disorder character | ized by a malformed, lateral curvatu | re of the spine. | I | 1 | |
| Soft tissue necrosis lower limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | zed by a necrotic process occurring | in the soft tissues of the lower ex | ctremity. | | |
| Soft tissue necrosis upper limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap | Life-threatening consequences; urgent intervention indicated | Death |

| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characterize | ed by fibrotic degeneration of the s | superficial soft tissues. | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, soft foods or purees | Decreased ROM with inability to adequately aliment or hydrate orally | - | - |
| Definition: A disorder characterize | ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | mastication. | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - 5 cm; shoe lift indicated; limiting instrumental ADL | , , | - | - |
| Definition: A disorder characterize | ed by of a discrepancy between th | e lengths of the lower or upper ex | tremities. | | |
| Musculoskeletal and connective tissue disorder - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Neoplasms benig | n, malignant and unspec | cified (incl cysts and poly | yps) | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Leukemia secondary to oncology chemotherapy | - | - | - | Present | Death |
| Definition: A disorder characterize | ed by leukemia arising as a result | of the mutagenic effect of chemot | herapy agents. | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by insufficiently healthy hemata | poietic cell production by the bone | e marrow. | | |
| Treatment related secondary malignancy | - | - | Non life-threatening secondary malignancy | Acute life-threatening secondary malignancy; blast crisis in leukemia | Death |
| Definition: A disorder characterize | ed by development of a malignanc | y most probably as a result of trea | atment for a previously existing ma | alignancy. | • |
| Tumor pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort from a ne | eoplasm that may be pressing on | a nerve, blocking blood vessels, ir | nflamed or fractured from metastas | sis. |
| Neoplasms benign, malignant<br>and unspecified (incl cysts and<br>polyps) - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Adverse Event Abducens nerve disorder Asymptomatic; clinical or diagnostic observations only; instrumental ADL instrumental A | care ADL limiting Severe symptoms; limiting self care ADL all nerve). limiting Severe symptoms; limiting self care ADL Severe symptoms; limiting self care ADL erve). So Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. memory self care ADL Voicelessness; unable to speak - - Voicelessness; unable to speak - - he vocal cords or may be functional (psychogenic). limiting Severe symptoms; limiting self care ADL Life-threatening consequences; urgent intervention indicated cent subarachnoid space. |
|---|---|
| Abducens nerve disorder Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the abducens nerve (sixth cranial nervection not indicated) Accessory nerve disorder Asymptomatic; clinical or diagnostic observations only; instrumental ADL instrumental ADL Definition: A disorder characterized by involvement of the accessory nerve (eleventh cranial nervection not indicated) Definition: A disorder characterized by involvement of the accessory nerve (eleventh cranial nervection not indicated) Definition: A disorder characterized by involvement of the accessory nerve (eleventh cranial nervection) not indicated Definition: A disorder characterized by involvement of the accustic nerve (eighth cranial nervectivity) Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and motor activity instrumental ADL Definition: A disorder characterized by systematic and extensive loss of memory. Definition: A disorder characterized by the inability to speak. It may result from injuries to the diagnostic observations only; instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact Ataxia Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by lack of coordination of muscle movements resulting Brachial plexopathy Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system As | limiting Severe symptoms; limiting self care ADL |
| diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the abducens nerve (sixth cranial nervention) and instrumental ADL Accessory nerve disorder Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the accessory nerve (eleventh cranial nervention) and indicated Definition: A disorder characterized by involvement of the accessory nerve (eleventh cranial nervention) and indicated of diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the accustic nerve (eighth cranial nervention) and indicated Definition: A disorder characterized by involvement of the accustic nerve (eighth cranial nervention) and indicated Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and Moderate; short term in loss; limiting instrument Definition: A disorder characterized by systematic and extensive loss of memory. Aphonia Definition: A disorder characterized by the inability to speak. It may result from injuries to the Arachnoiditis Mild symptoms Moderate symptoms; Instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact diagnostic observations only; instrumental ADL Definition: A disorder characterized by lack of coordination of muscle movements resulting Brachial plexopathy Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by a necrotic process occurring in the | care ADL limiting Severe symptoms; limiting self care ADL al nerve). limiting Severe symptoms; limiting self care ADL Severe symptoms; limiting self care ADL erve). s or Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. memory self care ADL Voicelessness; unable to speak - - Voicelessness; unable to speak - - he vocal cords or may be functional (psychogenic). limiting Severe symptoms; limiting self care ADL Cent subarachnoid space. limiting Severe symptoms; limiting self - - |
| Accessory nerve disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by involvement of the accessory nerve (eleventh cranic diagnostic observations only; instrumental ADL Accoustic nerve disorder NOS Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the accoustic nerve (eighth cranial new Moderate symptoms; linistrumental ADL Definition: A disorder characterized by involvement of the accoustic nerve (eighth cranial new Moderate restlessness increased motor activity instrumental ADL Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and Moderate; short term in loss; limiting instrumental ADL Definition: A disorder characterized by systematic and extensive loss of memory. Definition: A disorder characterized by the inability to speak. It may result from injuries to the Arachnoiditis Mild symptoms Moderate symptoms; linistrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjace Ataxia Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by lack of coordination of muscle movements resulting Moderate symptoms; linistrumental ADL Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regiona | Severe symptoms; limiting self care ADL all nerve). Ilimiting Severe symptoms; limiting self care ADL Severe symptoms; limiting self care ADL Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. Memory Ilimiting self care ADL Voicelessness; unable to speak |
| diagnostic observations only; intervential ADL Definition: A disorder characterized by involvement of the accessory nerve (eleventh crani diagnostic observations only; intervential ADL Definition: A disorder characterized by involvement of the accessory nerve (eleventh crani diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the acoustic nerve (eighth cranial new Moderate restlessness increased motor activity instrumental ADL Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and Moderate; short term in loss; limiting instrumental ADL Definition: A disorder characterized by systematic and extensive loss of memory. Definition: A disorder characterized by the inability to speak. It may result from injuries to the Arachnoiditis Mild symptoms Moderate symptoms; I instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact that is a disorder characterized by lack of coordination of muscle movements resulting Brachial plexopathy Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regional paresthesia of | care ADL all nerve). limiting Severe symptoms; limiting self care ADL erve). s or Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. memory Initian ADL Severe; long term memory loss; limiting self care ADL Voicelessness; unable to speak |
| Acoustic nerve disorder NOS Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the acoustic nerve (eighth cranial nerve that instrumental ADL Mild restlessness or increased motor activity instrumental ADL Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and Moderate; short term of loss; limiting instrumental ADL Definition: A disorder characterized by systematic and extensive loss of memory. Aphonia Definition: A disorder characterized by the inability to speak. It may result from injuries to the moderate symptoms; Instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact and adja | Severe symptoms; limiting self care ADL Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. Memory Initian ADL Voicelessness; unable to speak - - Voicelessness; unable to speak - - Noicelessness; unable to speak - - Voicelessness; unable to speak - - Severe symptoms; limiting self care ADL Life-threatening consequences; urgent intervention indicated Cent subarachnoid space. Limiting Severe symptoms; limiting self - - |
| diagnostic observations only; instrumental ADL Definition: A disorder characterized by involvement of the acoustic nerve (eighth cranial nerve) (high the properties) and the properties of the acoustic nerve (eighth cranial nerve) (high the properties) (high the p | care ADL so or Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. memory Severe; long term memory loss; limiting self care ADL Voicelessness; unable to speak |
| Mild restlessness or increased motor activity Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and Mild; transient memory loss Moderate; short term r loss; limiting instrument Poefinition: A disorder characterized by systematic and extensive loss of memory. Aphonia Definition: A disorder characterized by the inability to speak. It may result from injuries to the Arachnoiditis Mild symptoms Moderate symptoms; I instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact diagnostic observations only; intervention not indicated Definition: A disorder characterized by lack of coordination of muscle movements resulting diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | Severe restlessness or increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. Severe; long term memory loss; limiting self care ADL |
| motor activity increased motor activity increased motor activity instrumental ADL Definition: A disorder characterized by an uncomfortable feeling of inner restlessness and Moderate; short term reloss; limiting instrumental ADL Definition: A disorder characterized by systematic and extensive loss of memory. Aphonia | ty; limiting increased motor activity; limiting self care ADL inability to stay still; this is a side effect of some psychotropic drugs. Severe; long term memory loss; limiting self care ADL |
| Amnesia Mild; transient memory loss Moderate; short term reloss; limiting instrumer Definition: A disorder characterized by systematic and extensive loss of memory. Aphonia | Severe; long term memory loss; - - |
| Definition: A disorder characterized by systematic and extensive loss of memory. Aphonia Definition: A disorder characterized by the inability to speak. It may result from injuries to the symptoms; I instrumental ADL. Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact Ataxia Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by lack of coordination of muscle movements resulting Brachial plexopathy Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Moderate symptoms; orticosteroids indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | Voicelessness; unable to speak - - |
| Aphonia Definition: A disorder characterized by the inability to speak. It may result from injuries to the Arachnoiditis Mild symptoms Moderate symptoms; Instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjact and the arachnoid membrane and ad | he vocal cords or may be functional (psychogenic). Ilmiting Severe symptoms; limiting self care ADL Severe symptoms; limiting self urgent intervention indicated self severe symptoms; limiting self |
| Definition: A disorder characterized by the inability to speak. It may result from injuries to the Arachnoiditis Mild symptoms Moderate symptoms; Instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjace Ataxia Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by lack of coordination of muscle movements resulting and adjaced and adjaced are symptoms; Instrumental ADL Definition: A disorder characterized by lack of coordination of muscle movements resulting and Moderate symptoms; Instrumental ADL instrumental ADL instrumental ADL Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked and Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | he vocal cords or may be functional (psychogenic). Ilmiting Severe symptoms; limiting self care ADL Severe symptoms; limiting self urgent intervention indicated self severe symptoms; limiting self |
| Arachnoiditis Mild symptoms Moderate symptoms; I instrumental ADL Definition: A disorder characterized by inflammation of the arachnoid membrane and adjace Ataxia Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by lack of coordination of muscle movements resulting Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | limiting Severe symptoms; limiting self care ADL Severe symptoms; limiting self care ADL sent subarachnoid space. Severe symptoms; limiting self |
| Definition: A disorder characterized by inflammation of the arachnoid membrane and adjace Ataxia Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by lack of coordination of muscle movements resulting Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | cent subarachnoid space. limiting Severe symptoms; limiting self |
| Ataxia Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by lack of coordination of muscle movements resulting diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Moderate symptoms; corticosteroids indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | limiting Severe symptoms; limiting self |
| diagnostic observations only; instrumental ADL Definition: A disorder characterized by lack of coordination of muscle movements resulting Brachial plexopathy Asymptomatic; clinical or diagnostic observations only; instrumental ADL Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | |
| Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Asymptomatic; clinical or Moderate symptoms; observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | assistance indicated |
| diagnostic observations only; instrumental ADL Definition: A disorder characterized by regional paresthesia of the brachial plexus, marked Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | in the impairment or inability to perform voluntary activities. |
| Central nervous system Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | limiting Severe symptoms; limiting self care ADL - |
| diagnostic observations only; corticosteroids indicate intervention not indicated Definition: A disorder characterized by a necrotic process occurring in the brain and/or spin | discomfort and muscle weakness, and limited movement in the arm or hand. |
| | Severe symptoms; medical intervention indicated Life-threatening consequences; urgent intervention indicated |
| Derebrospinal fluid leakage Post-craniotomy: asymptomatic; Post-craniotomy: mod | nal cord. |
| Post-lumbar puncture: transient headache; postural care indicated; Post-lumbar puncture: persistent m symptoms; blood patcindicated | tervention indicated urgent intervention indicated report intervention indicated urgent indicated urgent indicated urg |
| Definition: A disorder characterized by loss of cerebrospinal fluid into the surrounding tissu | ies. |
| Cognitive disturbance Mild cognitive disability; not interfering with work/school/life performance; specialized educational services/devices not indicated Moderate cognitive dis interfering with work/sr performance but capal independent living; specialized resources on part time indicated | chool/life significant impairment of ble of work/school/life performance ecialized |
| Definition: A disorder characterized by a conspicuous change in cognitive function. | |
| Concentration impairment Mild inattention or decreased level of concentration attention or decreased concentration; limiting instrumental ADL | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Advance Event | 4 | | | 4 | |
| Adverse Event | Decrees distributed of slowly and | 2 | Difficult to arouse | | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to stimuli; limiting instrumental ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder characte | rized by a decrease in ability to perc | eive and respond. | • | • | |
| Dizziness | Mild unsteadiness or sensation | Moderate unsteadiness or | Severe unsteadiness or | - | - |
| | of movement | sensation of movement; limiting instrumental ADL | sensation of movement; limiting self care ADL | | |
| Definition: A disorder characte | rized by a disturbing sensation of lig | htheadedness, unsteadiness, gidd | liness, spinning or rocking. | | |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characte | rized by slow and slurred speech re | sulting from an inability to coordina | te the muscles used in speech. | | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Definition: A disorder characte | rized by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation. | | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet (e.g., oral supplements); noxious or unpleasant taste; loss of taste | - | - | - |
| Definition: A disorder characte | rized by abnormal sensual experien | ince with the taste of foodstuffs; it ca | n be related to a decrease in the s | sense of smell. | 1 |
| Dysphasia | Awareness of receptive or expressive characteristics; not impairing ability to communicate | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | - | - |
| Definition: A disorder characte | rized by impairment of verbal comm | unication skills, often resulting fron | n brain damage. | <del></del> | 1 |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | - |
| Definition: A disorder characte | rized by swelling due to an excessiv | e accumulation of fluid in the brain | l.<br>T | T | |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a pathologic process involving | ng the brain. | 1 | Г | |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary<br>movements; limiting<br>instrumental ADL | Severe involuntary movements or torticollis; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by abnormal, repetitive, involu | ntary muscle movements, frenzied | speech and extreme restlessness | S. | |
| Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a reduction in the strength of | of the facial muscles. | , | _ | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by involvement of the facial ne | rve (seventh cranial nerve). | | | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by involvement of the glossoph | naryngeal nerve (ninth cranial nerv | e). | | |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in various parts of the head | , not confined to the area of distrib | ution of any nerve. | |
| Hydrocephalus | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; intervention not indicated | Severe symptoms or neurological deficit; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal increase of ce | rebrospinal fluid in the ventricles o | f the brain. | ·<br> | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | - | - |
| Deficition: A disconder observator | rized by characterized by excessive | | • | • | • |

| | T | Nervous system dis | orucis | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the hypoglos | sal nerve (twelfth cranial nerve). | 1 | 1 | ' |
| Intracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the cranium. | | Intervention indicated | I | ı |
| Ischemia cerebrovascular | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | - | - | - |
| Definition: A disorder characteriz<br>damage. | ed by a decrease or absence of bl | ood supply to the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | ological |
| IVth nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the trochlear | nerve (fourth cranial nerve). | 1 | | |
| Lethargy | Mild symptoms; reduced alertness and awareness | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A disorder characteriz | ed by a decrease in consciousnes | s characterized by mental and ph | ysical inertness. | | |
| Leukoencephalopathy | Asymptomatic; small focal T2/FLAIR hyperintensities; involving periventricular white matter or <1/3 of susceptible areas of cerebrum +/- mild increase in subarachnoid space (SAS) and/or mild ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/3 to 2/3 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate ventriculomegaly | +/- moderate to severe increase | Life-threatening consequences; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Death |
| Definition: A disorder characteriz | ed by diffuse reactive astrocytosis | with multiple areas of necrotic for | i without inflammation. | | |
| Memory impairment | Mild memory impairment | Moderate memory impairment;<br>limiting instrumental ADL | Severe memory impairment;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a deterioration in memory fu | nction. | | | |
| Meningismus | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by neck stiffness, headache, ar | nd photophobia resulting from irrita | ation of the cerebral meninges. | | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by uncontrolled and purposeles | ss movements. | 1 | T | |
| Myelitis | Asymptomatic; mild signs (e.g., Babinski's reflex or Lhermitte's sign) | Moderate weakness or sensory loss; limiting instrumental ADL | Severe weakness or sensory loss; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the s | pinal cord. Symptoms include wea | akness, paresthesia, sensory loss, | marked discomfort and incontiner | nce. |
| Neuralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | red by intense painful sensation ald | ong a nerve or group of nerves. | | T | |
| Nystagmus | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involuntary movements of th | ie eyeballs. | T | T | |
| Oculomotor nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the oculomot | or nerve (third cranial nerve). | • | • | • |
| Olfactory nerve disorder | - | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | · | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz are experienced in the absence of | | ensory neurons resulting in abnorr | mal cutaneous sensations of tinglin | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneration | n of the peripheral motor nerves. | | | |
| Peripheral sensory neuropathy | Asymptomatic; loss of deep tendon reflexes or paresthesia | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | | n of the peripheral sensory nerves | | | |
| Phantom pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort related to | | ed from or is not physically part of | the body. | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| Definition: A disorder characteriz | ed by an episode of lightheadedne | ess and dizziness which may prec | ede an episode of syncope. | T | |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by dysfunction of the corticospi<br>nd a decrease in fine motor coord | | l cord. Symptoms include an incre | ease in the muscle tone in the lower | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting instrumental ADL; medical intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz connecting nerve root. | ed by inflammation involving a ner | ve root. Patients experience mark | ed discomfort radiating along a ne | erve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by paralysis of the recurrent lar | yngeal nerve. | | | |
| Reversible posterior leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very abnormal imaging studies; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | - | _ | | indings of posterior leukoencepha<br>s an acute or subacute reversible o | |
| Seizure | Brief partial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characteriz | ed by a sudden, involuntary skelet | tal muscular contractions of cerebi | ral or brain stem origin. | T | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort in the fac | ce, between the eyes, or upper tee | eth originating from the sinuses. | T | |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by characterized by excessive | sleepiness and drowsiness. | T | T | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle<br>tone and increase in resistance<br>through range of motion | Severe increase in muscle tone and increase in resistance through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characteriz disturbances. | ed by increased involuntary muscl | e tone that affects the regions inte | | It results in gait, movement, and s | peech |
| Stroke | Asymptomatic or mild neurologic deficit; radiographic findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a sudden loss of sensory fu | nction due to an intracranial vascu | lar event. | | + |
| Syncope Definition: A disorder characteriz | -<br>ed by spontaneous loss of conscio | <br> -<br>pusness caused by insufficient blo | Fainting; orthostatic collapse od supply to the brain. | - | - |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with or without imaging confirmation | - | - | - |
| Definition: A disorder characterize | ed by a brief attack (less than 24 h | nours) of cerebral dysfunction of va | ascular origin, with no persistent n | eurological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by the uncontrolled shaking mo | evement of the whole body or indiv | ridual parts. | | |
| Trigeminal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by involvement of the trigemina | al nerve (fifth cranial nerve). | | | |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by involvement of the vagus ne | rve (tenth cranial nerve). | • | | |
| Vasovagal reaction | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize increase in the stimulation of the | ed by a sudden drop of the blood progression vagus nerve. | pressure, bradycardia, and periph | eral vasodilation that may lead to | loss of consciousness. It results fr | om an |
| Nervous system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Pregna | ancy, puerperium and pe | rinatal conditions | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Fetal death | - | - | - | - | Fetal loss at<br>any<br>gestational<br>age |
| Definition: A disorder characterize | ed by death in utero; failure of the | product of conception to show evi | dence of respiration, heartbeat, or | definite movement of a voluntary | muscle after |
| expulsion from the uterus, without | t possibility of resuscitation. | | | | |
| Fetal growth retardation | - | <10% percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | - |
| Definition: A disorder characterize | ed by inhibition of fetal growth resu | ulting in the inability of the fetus to | achieve its potential weight. | | |
| Premature delivery | · | Delivery of a liveborn infant at >28 to 34 weeks gestation | Delivery of a liveborn infant at 24 to 28 weeks gestation | Delivery of a liveborn infant at 24 weeks of gestation or less | - |
| Definition: A disorder characterize gestation. | ed by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | tween the twentieth and thirty-sev | enth week of |
| Unintended pregnancy | - | - | Unintended pregnancy | - | - |
| Definition: A disorder characterize | ed by an unexpected pregnancy a | t the time of conception. | | • | • |
| Pregnancy, puerperium and perinatal conditions - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| | | Psychiatric disor | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | not indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by a state of restlessness asso | | Irritability and tension. | | |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by an inability to achieve orgas | | | 1 | 1 |
| Anxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization not indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder characte stimulus. | erized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dys | pnea unattached to a clearly iden | tifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by a lack of clear and orderly the | nought and behavior. | 1 | 1 | Г |
| Delayed orgasm | Delay in achieving orgasm not adversely affecting relationship | Delay in achieving orgasm adversely affecting relationship | - | - | - |
| | erized by sexual dysfunction characte | | 1. | | 1 |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder character<br>reversible condition. | erized by the acute and sudden devel | opment of confusion, illusions, mo | ovement changes, inattentiveness, | agitation, and hallucinations. Usu | ally, it is a |
| | | Moderate delucional symptoms | Sovere delucional aymptoma: | Life threatening consequences | Dooth |
| Delusions | - | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by false personal beliefs held o | ontrary to reality, despite contradi | ctory evidence and common sens | e. | 1 |
| Depression | Mild depressive symptoms | Moderate depressive symptoms; limiting instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by melancholic feelings of grief | or unhappiness. | | | |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | - |
| Definition: A disorder characte | erized by an exaggerated feeling of w | ell-being which is disproportionate | to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by a false sensory perception in | n the absence of an external stime | ulus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling<br>asleep, staying asleep or<br>waking up early | - | - |
| Definition: A disorder characte | erized by difficulty in falling asleep and | d/or remaining asleep. | | | |
| Libido decreased | Decrease in sexual interest not adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by a decrease in sexual desire | T | T | T | 1 |
| Libido increased | Mild increase in sexual interest not adversely affecting relationship | Moderate increase in sexual interest adversely affecting relationship | Severe increase in sexual interest leading to dangerous behavior | - | - |
| Definition: A disorder characte | erized by an increase in sexual desire | ·<br>· | • | • | • |
| Mania | Mild manic symptoms (e.g., elevated mood, rapid thoughts, rapid speech, decreased need for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g., hypomania; major sexual or financial indiscretions); hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by excitement of psychotic prop | portions manifested by mental and | d physical hyperactivity, disorganiz | ation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |

| | | Psychiatric disord | ders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by a conspicuous change in a p | person's behavior and thinking. | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characterize tumor. | ed by personality change, impaired | d functioning, and loss of touch wi | th reality. It may be a manifestatio | n of schizophrenia, bipolar disorde | er or brain |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an inability to rest, relax or b | pe still. | | | |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide<br>with serious intent to die which<br>requires hospitalization | - |
| Definition: A disorder characterize | ed by thoughts of taking one's owr | n life. | | | |
| Suicide attempt | - | - | Suicide attempt or gesture<br>without intent to die which may<br>not require hospitalization | Suicide attempt with intent to die which requires hospitalization | Death |
| Definition: A disorder characterize | ed by self-inflicted harm in an atter | mpt to end one's own life. | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |

| Renal and urinary disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute kidney injury Definition: A disorder character | Creatinine level increase of >0.3 mg/dL; creatinine 1.5 - 2.0 x above baseline ized by the acute loss of renal functions. | baseline | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated | Life-threatening consequences; dialysis indicated | Death |
| causes (ureteral or bladder out | • | , | | ,,, | |
| Bladder perforation | - | Extraperitoneal perforation, indwelling catheter indicated | Intraperitoneal perforation;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>organ failure; urgent operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by a rupture in the bladder wall | | 1 | <u> </u> | |
| Bladder spasm | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | - | - |
| Definition: A disorder character | ized by a sudden and involuntary co | ontraction of the bladder wall. | | | |
| Chronic kidney disease | eGFR (estimated Glomerular<br>Filtration Rate) or CrCl<br>(creatinine clearance) <lln -="" 60<br="">ml/min/1.73 m2 or proteinuria<br/>2+ present; urine<br/>protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated | Death |
| Definition: A disorder character | ized by gradual and usually perman | ent loss of kidney function resulting | ng in renal failure. | <b>-</b> | |
| Cystitis noninfective | Microscopic hematuria; minimal increase in frequency, urgency, dysuria, or nocturia; new onset of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the bladder | ,<br>which is not caused by an infectio | n of the urinary tract. | • | |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self care ADL | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate blood in the urine. | | | |
| Hemoglobinuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate the presence of free hemo | globin in the urine. | | |
| Proteinuria | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 - 3.4 g/24 hrs;<br>Pediatric: urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5<br>g/24 hrs;<br>Pediatric: urine P/C >1.9 | - | - |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate the presence of excessive | protein in the urine. It is predomin | antly albumin, but also globulin. | |
| Renal calculi | Asymptomatic or mild<br>symptoms; occasional use of<br>nonprescription analgesics<br>indicated | Symptomatic; oral antiemetics indicated; around the clock nonprescription analgesics or any oral narcotic analgesics indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences;<br>urgent radiologic, endoscopic or<br>operative intervention indicated | Death |
| Definition: A disorder character | ized by the formation of crystals in t | he pelvis of the kidney. | | <u> </u> | 1 |
| Renal colic | Mild pain not interfering with activity; nonprescription medication indicated | Moderate pain; limiting instrumental ADL; prescription medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |

| | | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or<br>hospitalization indicated;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | rized by bleeding from the kidney. | | | | |
| Urinary fistula | - | Noninvasive intervention indicated; urinary or suprapubic catheter placement indicated | Limiting self care ADL; elective<br>radiologic, endoscopic or<br>operative intervention indicated;<br>permanent urinary diversion<br>indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between any part of the urinary s | system and another organ or anato | omic site. | |
| Urinary frequency | Present | Limiting instrumental ADL; medical management indicated | - | - | - |
| Definition: A disorder character | rized by urination at short intervals. | T | T | T | |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder character | rized by inability to control the flow o | f urine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by accumulation of urine within | the bladder because of the inabil | ity to urinate. | | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by blockage of the normal flow | of contents of the urinary tract. | , | T | |
| Urinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | omfort in the urinary tract. | 1 | | |
| Urinary urgency | Present | Limiting instrumental ADL;<br>medical management indicated | - | - | - |
| Definition: A disorder character | rized by a sudden compelling urge to | urinate. | _ | T | |
| Jrine discoloration | Present | - | - | - | - |
| Definition: A disorder character | rized by a change in the color of the | urine. | | | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azoospermia | - | - | Absence of sperm in ejaculate | - | - |
| Definition: A disorder characte | erized by laboratory test results that in | ndicate complete absence of speri | matozoa in the semen. | | |
| Breast atrophy | Minimal asymmetry; minimal | Moderate asymmetry; moderate | Asymmetry >1/3 of breast | - | - |
| . , | atrophy | atrophy | volume; severe atrophy | | |
| Definition: A disorder characte | erized by underdevelopment of the br | east. | ' | ' | • |
| Breast pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | _ |
| , | · | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by marked discomfort sensatio | n in the breast region. | ' | ' | • |
| Dysmenorrhea | Mild symptoms; intervention not | | Severe symptoms; limiting self | _ | _ |
| _, | indicated | instrumental ADL | care ADL | | |
| Definition: A disorder characte | rized by abnormally painful abdomin | al cramps during menses. | ! | ! | ' |
| Dyspareunia | Mild discomfort or pain | Moderate discomfort or pain | Severe discomfort or pain | | _ |
| 3y3parcuma | associated with vaginal | associated with vaginal | associated with vaginal | | |
| | penetration; discomfort relieved | penetration; discomfort or pain | penetration; discomfort or pain | | |
| | with use of vaginal lubricants or | partially relieved with use of | unrelieved by vaginal lubricants | | |
| | estrogen | vaginal lubricants or estrogen | or estrogen | | |
| Definition: A disorder characte | erized by painful or difficult coitus. | | | | |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde | - | - | - |
| | | ejaculation | | | |
| Definition: A disorder characte | erized by problems related to ejaculat | ion. This category includes prema | ture, delayed, retrograde and pair | ful ejaculation. | • |
| Erectile dysfunction | Decrease in erectile function | Decrease in erectile function | Decrease in erectile function | - | _ |
| | (frequency or rigidity of | (frequency/rigidity of erections), | (frequency/rigidity of erections) | | |
| | erections) but intervention not | erectile intervention indicated, | but erectile intervention not | | |
| | indicated (e.g., medication or | (e.g., medication or mechanical | helpful (e.g., medication or | | |
| | use of mechanical device, | devices such as penile pump) | mechanical devices such as | | |
| | penile pump) | | penile pump); placement of a | | |
| | | | permanent penile prosthesis | | |
| | | | indicated (not previously | | |
| 5 5 W A F A F A F | | | present) | | I |
| | erized by the persistent or recurrent in | | | | T |
| Fallopian tube obstruction | Diagnostic observations only; | Mild symptoms; elective | Severe symptoms; elective | - | - |
| | intervention not indicated | intervention indicated | operative intervention indicated | ļ | I |
| Definition: A disorder characte | erized by blockage of the normal flow | of the contents in the fallopian tub | oe. | | |
| Fallopian tube stenosis | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| | diagnostic observations only; | not indicated | operative intervention indicated | urgent operative intervention | |
| | intervention not indicated | | | indicated (e.g., organ resection) | |
| Definition: A disorder characte | erized by a narrowing of the fallopian | tube lumen. | ī | 1 | |
| Female genital tract fistula | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| | diagnostic observations only; | not indicated | operative intervention indicated | urgent intervention indicated | |
| | intervention not indicated | | | | |
| Definition: A disorder characte | erized by an abnormal communication | between a female reproductive s | ystem organ and another organ o | r anatomic site. | |
| Feminization acquired | Mild symptoms; intervention not | Moderate symptoms; medical | - | - | - |
| | indicated | intervention indicated | | | |
| Definition: A disorder characte | erized by the development of seconda | ary female sex characteristics in m | nales due to extrinsic factors. | | _ |
| Genital edema | Mild swelling or obscuration of | Readily apparent obscuration of | Lymphorrhea; gross deviation | - | - |
| | anatomic architecture on close | anatomic architecture; | from normal anatomic contour; | | |
| | inspection | obliteration of skin folds; readily | limiting self care ADL | | |
| | | apparent deviation from normal | | | |
| | | anatomic contour | | | I |
| Definition: A disorder characte | erized by swelling due to an excessive | e accumulation of fluid in the genit | als. | 1 | |
| Gynecomastia | Asymptomatic breast | Symptomatic (e.g., pain or | Severe symptoms; elective | - | - |
| | enlargement | psychosocial impact) | operative intervention indicated | | |
| Definition: A disorder characte | erized by excessive development of the | ne breasts in males. | | | |
| -lematosalpinx | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| • | imaging study or laparoscopy; | intervention indicated | indicated; radiologic or | urgent operative intervention | |
| | intervention not indicated | | endoscopic intervention | indicated | |

| ormally heavy vaginal bl<br>matic; asymmetry with<br>action and/or<br>g of the nipple areolar<br>alformation of the nipple<br>incentration >48<br>or motility >68% | Intermittent menses with skipped menses for more than 4 to 6 months menses. Changes in lactation, significantly affecting breast production or expression of breast milk on. It is not necessarily related to p. Moderate symptoms; medical intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex | Grade 3 Persistent amenorrhea for more than 6 months - pregnancy that is observed in female services in the service of the services of the | - ales and can be observed in males Life-threatening consequences; urgent intervention indicated | - Death |
|---|---|---|---|---|
| presence of blood in a fant menses with menses for no more 3 months ular cycle or duration of ges in lactation, not the action of breast milk surbances of milk secretic supplements indicated promally heavy vaginal bloomatic; asymmetry with action and/or g of the nipple arcentration >48 or motility >68% crease in the number of | Intermittent menses with skipped menses for more than 4 to 6 months femenses. Changes in lactation, significantly affecting breast production or expression of breast milk on. It is not necessarily related to p. Moderate symptoms; medical intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Persistent amenorrhea for more than 6 months - pregnancy that is observed in female Severe; transfusion indicated; surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | - ales and can be observed in males | - |
| nt menses with nenses for no more 3 months ular cycle or duration of ges in lactation, not tly affecting production sion of breast milk urbances of milk secretic supplements indicated ormally heavy vaginal bl matic; asymmetry with action and/or g of the nipple areolar ulafformation of the nipple mentration >48 or motility >68% crease in the number of | Intermittent menses with skipped menses for more than 4 to 6 months in menses. Changes in lactation, significantly affecting breast production or expression of breast milk on. It is not necessarily related to publicate milk on the intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | than 6 months - pregnancy that is observed in female Severe; transfusion indicated; surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | Life-threatening consequences; | |
| nenses for no more 3 months ular cycle or duration of ges in lactation, not tity affecting production sion of breast milk urbances of milk secretic supplements indicated ormally heavy vaginal bl matic; asymmetry with action and/or g of the nipple areolar alformation of the nipple incentration >48 or motility >68% crease in the number of | skipped menses for more than 4 to 6 months for menses. Changes in lactation, significantly affecting breast production or expression of breast milk on. It is not necessarily related to publicate more more more more more more more mor | than 6 months - pregnancy that is observed in female Severe; transfusion indicated; surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | Life-threatening consequences; | |
| ges in lactation, not tly affecting production sion of breast milk urbances of milk secretic supplements indicated ormally heavy vaginal bl matic; asymmetry with action and/or g of the nipple areolar alformation of the nipple uncentration >48 or motility >68% crease in the number of | Changes in lactation, significantly affecting breast production or expression of breast milk on. It is not necessarily related to pure moderate symptoms; medical intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Severe; transfusion indicated; surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | Life-threatening consequences; | |
| tly affecting production sion of breast milk scretch supplements indicated supplements as a supplement of the nipple area of the nipple supplement of the nipple supplement of the nipple supplement of the nipplement of the nipplement of the number of the nu | significantly affecting breast production or expression of breast milk on. It is not necessarily related to p Moderate symptoms; medical intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Severe; transfusion indicated; surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | Life-threatening consequences; | |
| ormally heavy vaginal bl<br>matic; asymmetry with<br>action and/or<br>g of the nipple areolar<br>alformation of the nipple<br>encentration >48<br>or motility >68%<br>crease in the number of | Moderate symptoms; medical intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Severe; transfusion indicated; surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | Life-threatening consequences; | |
| ormally heavy vaginal bl<br>matic; asymmetry with<br>action and/or<br>g of the nipple areolar<br>alformation of the nipple<br>oncentration >48<br>- or motility >68%<br>crease in the number of | intervention indicated (e.g., hormones) eeding during menses. Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | surgical intervention indicated (e.g., hysterectomy) - Sperm concentration <13 | | Death - |
| natic; asymmetry with action and/or g of the nipple areolar alformation of the nipple oncentration >48 and or motility >68% crease in the number of | Symptomatic; asymmetry of nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | 1 ' | - | - |
| action and/or g of the nipple areolar alformation of the nipple uncentration >48 L or motility >68% crease in the number of | nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Sperm concentration 13 - 48 million/mL or motility 32 - 68% | 1 ' | - | - |
| ncentration >48<br>_ or motility >68%<br>crease in the number of | Sperm concentration 13 - 48 million/mL or motility 32 - 68% | 1 ' | - | |
| or motility >68%<br>crease in the number of | million/mL or motility 32 - 68% | 1 ' | - | |
| | spermatozoa in the semen. | | | - |
| leeding identified on | | 1 | | |
| tudy or laproscopy;<br>on not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| ding from the ovary. | I | ı | ı | ' |
| natic clinical or<br>c observations only;<br>on not indicated | Symptomatic and intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| ng or disruption of the o | varian tissue. | , | • | ' |
| | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| ked discomfort sensation | n in one side of the abdomen betw | veen menstrual cycles, around the | time of the discharge of the ovum | from the |
| natic; clinical or<br>c observations only;<br>on not indicated | Symptomatic, not interfering<br>with bladder, bowel, or vaginal<br>function; limiting instrumental<br>ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| duction in the strength o | f the muscles of the pelvic floor. | | | 1 |
| | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| ked discomfort sensation | n in the pelvis. | T | Γ | |
| | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| ked discomfort sensation | n in the penis. | Ī | <u> </u> | |
| | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | omfort in the area between the gen | ital organs and the anus. | Т | I |
| nsation of marked disco | - | Present | - | - |
| nsation of marked disco | | shes, night sweats, mood swings a<br>Severe bleeding; transfusion | Life-threatening consequences; urgent operative intervention | Death |
| (6 | sation of marked disco | instrumental ADL ed discomfort sensation in the penis. Moderate pain; limiting instrumental ADL sation of marked discomfort in the area between the ger | instrumental ADL ADL ad discomfort sensation in the penis. Moderate pain; limiting instrumental ADL ADL sation of marked discomfort in the area between the genital organs and the anus. - Present an failure before the age of 40. Symptoms include hot flashes, night sweats, mood swings are deding identified on udy; intervention not indicated intervention indicated Moderate bleeding; medical intervention indicated indicated; radiologic or | instrumental ADL ADL ad discomfort sensation in the penis. Moderate pain; limiting instrumental ADL ADL Moderate pain; limiting instrumental ADL ADL sation of marked discomfort in the area between the genital organs and the anus. - Present - an failure before the age of 40. Symptoms include hot flashes, night sweats, mood swings and a decrease in sex drive. Deeding identified on Moderate bleeding; medical Severe bleeding; transfusion Life-threatening consequences; |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | red by bleeding from the prostate of | pland. | 1 | | |
| Prostatic obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz<br>tream, and incomplete emptyin | zed by compression of the urethra | secondary to enlargement of the p | prostate gland. This results in voidi | ng difficulties (straining to void, sl | ow urine |
| Prostatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the prostate gland. | | | |
| Scrotal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the scrotal area. | <del>,</del> | | |
| Spermatic cord hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the spermatic | cord. | | | |
| Spermatic cord obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | red by blockage of the normal flow | of the contents of the spermatic c | ord. | | |
| Festicular disorder | Asymptomatic; clinical or diagnostic observations only; | Symptomatic but not interfering with urination or sexual | Severe symptoms; interfering with urination or sexual function; | Life-threatening consequences; urgent intervention indicated | Death |
| | intervention not indicated | activities; intervention not indicated; limiting instrumental ADL | limiting self care ADL;<br>intervention indicated | | |
| Definition: A disorder characteriz | zed by involvement of the testis. | I | 1 | I | ı |
| Testicular hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by bleeding from the testis. | 1 | 1 | | |
| esticular pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the testis. | | T | |
| Jterine fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | n between the uterus and another | organ or anatomic site. | I | 1 |
| Jterine hemorrhage | <u> </u> | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the uterus. | • | | • | |
| Iterine obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | zed by blockage of the uterine outle | et. | | | |
| Iterine pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| efinition: A disorder characteriz | red by a sensation of marked disco | omfort in the uterus. | 1 | | |
| 'aginal discharge | Mild vaginal discharge (greater than baseline for patient) | Moderate to heavy vaginal discharge; use of perineal pad or tampon indicated | - | - | - |
| Definition: A disorder characterize | ed by vaginal secretions. Mucus p | | discharged from the vagina natura | lly, especially during the childbea | ring years. |
| /aginal dryness | Mild vaginal dryness not interfering with sexual function | Moderate vaginal dryness interfering with sexual function | Severe vaginal dryness resulting in dyspareunia or | - | - |
| Definition: A disorder characteriz | l<br>red by an uncomfortable feeling of | or causing frequent discomfort itching and burning in the vagina. | severe discomfort | I | 1 |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between the vagina and another | organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on<br>clinical exam or imaging study;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema, or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal<br>ulceration; life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation involving the v | agina. Symptoms may include red | lness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characterize | ed by blockage of vaginal canal. | | 1 | | |
| Vaginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | mfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a rupture in the vaginal wall. | | | | • |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or shortening not interfering with physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characterize | ed by a narrowing of the vaginal c | anal. | | | |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | - | - |
| Definition: A disorder characterize intercourse. | ed by involuntary spasms of the po | elvic floor muscles, resulting in pa | thologic tightness of the vaginal w | all during penetration such as duri | ng sexual |
| Reproductive system and breast<br>disorders - Other, specify | * ' | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adult respiratory distress<br>syndrome | - | - | Present with radiologic findings; intubation not indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri<br>surgery. | zed by progressive and life-threater | ning pulmonary distress in the abs | ence of an underlying pulmonary | condition, usually following major t | rauma or |
| Allergic rhinitis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| | zed by an inflammation of the nasa<br>s of the sinuses, eyes, middle ear, a | • | • | • | ay also |
| Apnea | - | - | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by cessation of breathing. | I | I | T | |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Altered eating habits; coughing or choking episodes after eating or swallowing; medical intervention indicated (e.g., suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by inhalation of solids or liquids | s into the lungs. | | <u> </u> | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by the collapse of part or the e | ntire lung. | T | T | 1 |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | · | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild<br>wheezing); endoscopic<br>evaluation indicated;<br>radiographic evidence of<br>atelectasis/lobar collapse;<br>medical management indicated<br>(e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by blockage of a bronchus pas | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | zed by a narrowing of the bronchial | | | leg at the second | <b>.</b> |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between a bronchus and the ple | ural cavity. | T | ı |
| Bronchopulmonary hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g., | Life-threatening respiratory or hemodynamic compromise; intubation or urgent intervention | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bronchospasm | Mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Limiting self care ADL; oxygen saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a sudden contraction of the | smooth muscles of the bronchial | wall. | 1 | |
| Chylothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thoracentesis or tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | rized by milky pleural effusion (abno | rmal collection of fluid) resulting fr | om accumulation of lymph fluid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription intervention indicated | Moderate symptoms, medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte by a distinctive sound. | rized by sudden, often repetitive, spa | asmodic contraction of the thoraci | c cavity, resulting in violent release | e of air from the lungs and usually | accompani |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an uncomfortable sensation | of difficulty breathing. | | | , |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; topical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the nose. | 1 | | | |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe symptoms; interfering with sleep; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by repeated gulp sounds that re | esult from an involuntary opening | and closing of the glottis. This is a | attributed to a spasm of the diaphra | igm. |
| Hoarseness | Mild or intermittent voice change; fully understandable; self-resolves | Moderate or persistent voice<br>changes; may require<br>occasional repetition but<br>understandable on telephone;<br>medical evaluation indicated | Severe voice changes including predominantly whispered speech | - | - |
| Definition: A disorder characte | rized by harsh and raspy voice arisir | ng from or spreading to the larynx. | | | |
| Нурохіа | - | Decreased oxygen saturation<br>with exercise (e.g., pulse<br>oximeter <88%); intermittent<br>supplemental oxygen | Decreased oxygen saturation at<br>rest (e.g., pulse oximeter <88%<br>or PaO2 <=55 mm Hg) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | rized by a decrease in the level of ox | | 1. | 1 . | |
| Laryngeal edema | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | Stridor; respiratory distress;<br>hospitalization indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | rized by swelling due to an excessive | | 1 | | |
| _aryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characte | ा<br>rized by an abnormal communication | between the larynx and another | organ or anatomic site. | , | 1 |
| _aryngeal hemorrhage | Mild cough or trace hemoptysis; laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic, endoscopic, or operative intervention indicated (e.g., | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | | | hemostasis of bleeding site) | Intubation) | l |
| Definition: A disorder characte | rized by bleeding from the larynx. | | nemostasis of bleeding site) | Intubation) | |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngeal mucositis | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered oral intake | Severe pain; severely altered<br>eating/swallowing; medical<br>intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteri | ized by an inflammation involving th | e mucous membrane of the laryn | (. | i . | |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ized by blockage of the laryngeal ai | rway. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| | ized by a narrowing of the laryngea | | | | <b>.</b> |
| Laryngopharyngeal dysesthesia | a Mild symptoms; no anxiety;<br>intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and swallowing difficulty; limiting self care ADL | Life-threatening consequences | Death |
| Definition: A disorder characteri | ized by an uncomfortable persistent | sensation in the area of the laryn | gopharynx. | <b>-</b> | |
| Laryngospasm | - | Transient episode; intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characteri | ized by paroxysmal spasmodic mus | cular contraction of the vocal cord | | | ' |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hemostasis of bleeding<br>site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ized by bleeding from the mediastin | um. | 1 ' | l | 1 |
| Nasal congestion | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Associated with bloody nasal discharge or epistaxis | - | - |
| | ized by obstruction of the nasal pas | 1 | | 17.11 | n |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ized by an abnormal communication | n between the pharynx and anothe | er organ or anatomic site. | 1 | |
| Pharyngeal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | ized by bleeding from the pharynx. | | | | 1 |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics indicated; altered oral intake; limiting instrumental ADL | Severe pain; unable to adequately aliment or hydrate orally; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ized by an inflammation involving th | e mucous membrane of the phary | rnx. | Γ | ı |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Respi | ratory, thoracic and med | lastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | rized by a necrotic process occurring | in the pharynx. | <u> </u> | | |
| Pharyngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder character | rized by a narrowing of the pharynge | al airway. | , | • | • |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by marked discomfort sensation | n in the pharyngolaryngeal region. | | | |
| Pleural effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., diuretics or limited therapeutic thoracentesis) | Symptomatic with respiratory<br>distress and hypoxia; surgical<br>intervention including chest tube<br>or pleurodesis indicated | indicated | Death |
| Definition: A disorder character | rized by an increase in amounts of flo | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or associated with pneumothorax; chest tube drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | rized by bleeding from the pleural ca | vity. | • | | • |
| Pleuritic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by marked discomfort sensation | n in the pleura. | T | T | |
| Pneumonitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | rized by inflammation focally or diffus | | | | I |
| Pneumothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative intervention indicated; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by abnormal presence of air in | the pleural cavity resulting in the | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | rized by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | |
| Productive cough | | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | - | - |
| | rized by expectorated secretions upo | | | Life iii | L |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at rest; oxygen indicated; limiting self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder character | rized by accumulation of fluid in the I | ung tissues that causes a disturba | nce of the gas exchange that may | lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia; radiologic<br>pulmonary fibrosis <25% of lung<br>volume | Moderate hypoxemia; evidence<br>of pulmonary hypertension;<br>radiographic pulmonary fibrosis<br>25 - 50% | Severe hypoxemia; evidence of right-sided heart failure; radiographic pulmonary fibrosis >50 - 75% | Life-threatening consequences (e.g., hemodynamic/pulmonary complications); intubation with ventilatory support indicated; radiographic pulmonary fibrosis >75% with severe honeycombing | Death |
| Definition: A disorder character | rized by the replacement of the lung | tissue by connective tissue, leadir | ng to progressive dyspnea, respira | tory failure or right heart failure. | |
| Pulmonary fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Respi | ratory, thoracic and med | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | zed by an abnormal communication | | | ler u | <b>.</b> |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other | Moderate dyspnea, cough; requiring evaluation by cardiac | Severe symptoms, associated with hypoxemia, right heart | Life-threatening airway consequences; urgent | Death |
| | evaluation | catheterization and medical intervention | failure; oxygen indicated | intervention indicated (e.g., tracheotomy or intubation) | |
| Definition: A disorder characteri | zed by an increase in pressure with | nin the pulmonary circulation due to | lung or heart disorder. | | |
| Respiratory failure | - | - | - | Life-threatening consequences; urgent intervention, intubation, | Death |
| | | | | or ventilatory support indicated | |
| Definition: A disorder characteri<br>with an increase in arterial level | zed by impaired gas exchange by t | he respiratory system resulting in | hypoxemia and a decrease in oxy | genation of the tissues that may be | e associat |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight | Moderate signs or symptoms; | Severe symptoms; | Life-threatening consequences; | Death |
| Council asia synaromo | gain; intervention with fluid restriction and/or diuretics indicated | steroids indicated | hospitalization indicated | ventilatory support indicated | Boun |
| Definition: A disorder characteri | zed by weight gain, dyspnea, pleur | ।<br>al and pericardial effusions, leukoo | l<br>cytosis and/or renal failure original | I<br>ly described in patients treated wit | ।<br>th all-trans |
| Sinus disorder | Asymptomatic mucosal crusting; | | Stenosis with significant nasal | Necrosis of soft tissue or bone; | Death |
| | blood-tinged secretions | edema/narrowing interfering<br>with airflow; limiting instrumental<br>ADL | obstruction; limiting self care<br>ADL | urgent operative intervention indicated | |
| Definition: A disorder characteri | l<br>zed by involvement of the paranasa | 1 | | I | Į. |
| Sleep apnea | Snoring and nocturnal sleep | Moderate apnea and oxygen | Oxygen desaturation; | Cardiovascular or | Death |
| | arousal without apneic periods | desaturation; excessive daytime | associated with hypertension; | neuropsychiatric symptoms; | |
| | | sleepiness; medical evaluation indicated; limiting instrumental | medical intervention indicated;<br>limiting self care ADL | urgent operative intervention indicated | |
| Definition: A disorder characteri | <br>zed by cessation of breathing for sh | ADL | | | |
| Sneezing | Mild symptoms; intervention not | | - | - | - |
| 3 | indicated | intervention indicated | | | |
| Definition: A disorder characteri | zed by the involuntary expulsion of | air from the nose. | | | |
| Sore throat | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL; limiting ability to swallow | | |
| | zed by of marked discomfort in the | throat | | T . | |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention | Life-threatening airway compromise; urgent intervention | Death |
| | | | indicated | indicated (e.g., tracheotomy or | |
| | | | | intubation) | |
| Definition: A disorder characteri | zed by a high pitched breathing sou | und due to laryngeal or upper airw | ay obstruction. | T | |
| Tracheal fistula | Asymptomatic; clinical or | Symptomatic; tube | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | diagnostic observations only;<br>intervention not indicated | thoracostomy or medical intervention indicated; limiting | care ADL; endoscopic or operative intervention indicated | urgent operative intervention indicated (e.g., thoracoplasty, | |
| | intervention not maioatou | instrumental ADL | (e.g., stent or primary closure) | chronic open drainage or | |
| | | | | multiple thoracotomies) | |
| Definition: A disorder characteri | zed by an abnormal communication | between the trachea and anothe | organ or anatomic site. | · | |
| Tracheal mucositis | Endoscopic findings only; | Moderate symptoms; medical | Severe pain; hemorrhage or | Life-threatening consequences; | Death |
| | minimal hemoptysis, pain, or respiratory symptoms | intervention indicated; limiting instrumental ADL | respiratory symptoms; limiting self care ADL | urgent intervention indicated | |
| Definition: A disorder characteri | | 1 | | l | I |
| Definition: A disorder characteri.<br>Tracheal stenosis | zed by an inflammation involving th | | ea.<br>Stridor or respiratory distress | Life-threatening airway | Death |
| 114011041 310110313 | Asymptomatic; clinical or diagnostic observations only; | Symptomatic (e.g., noisy airway breathing), but causing no | limiting self care ADL; | compromise; urgent intervention | Deam |
| | intervention not indicated | respiratory distress; medical | endoscopic intervention | indicated (e.g., tracheotomy or | |
| | | management indicated (e.g., steroids) | indicated (e.g., stent, laser) | intubation) | |
| Definition: A disorder characteri | zed by a narrowing of the trachea. | | | | |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Voice alteration | Mild or intermittent change from normal voice | Moderate or persistent change<br>from normal voice; still<br>understandable | Severe voice changes including<br>predominantly whispered<br>speech; may require frequent<br>repetition or face-to-face contact<br>for understandability; may<br>require assistive technology | - | 1 |
| Definition: A disorder characterize | ed by a change in the sound and/o | or speed of the voice. | | | |
| Wheezing | Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe respiratory symptoms<br>limiting self care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a high-pitched, whistling sou | and during breathing. It results from | n the narrowing or obstruction of t | he respiratory airways. | |
| Respiratory, thoracic and mediastinal disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Alopecia | Hair loss of <50% of normal for<br>that individual that is not<br>obvious from a distance but only<br>on close inspection; a different<br>hair style may be required to | Hair loss of >=50% normal for<br>that individual that is readily<br>apparent to others; a wig or hair<br>piece is necessary if the patient<br>desires to completely | - | - | - |
| | cover the hair loss but it does<br>not require a wig or hair piece to<br>camouflage | camouflage the hair loss;<br>associated with psychosocial<br>impact | | | |
| Definition: A disorder characteri | zed by a decrease in density of hair | compared to normal for a given i | ndividual at a given age and body | location. | _ |
| Body odor | Mild odor; physician intervention not indicated; self care interventions | Pronounced odor; psychosocial impact; patient seeks medical intervention | - | - | - |
| Definition: A disorder characteri | zed by an abnormal body smell res | ulting from the growth of bacteria | on the body. | 1 | |
| Bullous dermatitis | Asymptomatic; blisters covering <10% BSA | Blisters covering 10 - 30% BSA;<br>painful blisters; limiting<br>instrumental ADL | Blisters covering >30% BSA;<br>limiting self care ADL | Blisters covering >30% BSA;<br>associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder characteri | zed by inflammation of the skin cha | racterized by the presence of bull | ae which are filled with fluid. | T | 1 |
| Dry skin | Covering <10% BSA and no associated erythema or pruritus | Covering 10 - 30% BSA and associated with erythema or pruritus; limiting instrumental ADL | Covering >30% BSA and associated with pruritus; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by flaky and dull skin; the pores | are generally fine, the texture is | a papery thin texture. | · | _ |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target lesions covering 10 -<br>30% BSA and associated with<br>skin tenderness | Target lesions covering >30%<br>BSA and associated with oral or<br>genital erosions | Target lesions covering >30%<br>BSA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder characteri | zed by target lesions (a pink-red rin | g around a pale center). | T | T | 1 |
| Erythroderma | - | Erythema covering >90% BSA without associated symptoms; limiting instrumental ADL | Erythema covering >90% BSA with associated symptoms (e.g., pruritus or tenderness); limiting self care ADL | Erythema covering >90% BSA with associated fluid or electrolyte abnormalities; ICU care or burn unit indicated | Death |
| Definition: A disorder characteri | zed by generalized inflammatory er | ythema and exfoliation. The inflan | nmatory process involves > 90% o | f the body surface area. | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL | Covering >30% BSA;<br>associated with erythema or<br>tenderness; limiting self-care<br>ADL | - | - |
| Definition: A disorder characteri | zed by shrinking of adipose tissue. | | T | T | 1 |
| Hirsutism | In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | - | - | - |
| Definition: A disorder characteri | zed by the presence of excess hair | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | and unde |
| androgen control (beard, moust | • • | | | | |
| Hyperhidrosis | Limited to one site (palms, soles, or axillae); self care interventions | Involving >1 site; patient seeks<br>medical intervention; associated<br>with psychosocial impact | Generalized involving sites<br>other than palms, soles, or<br>axillae; associated with<br>electrolyte/hemodynamic | - | - |

| | Sk | in and subcutaneous tis | sue alsoraers | | |
|---|---|---|---|---|---|
| | | I | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or<br>density of hair that the patient is<br>either able to camouflage by<br>periodic shaving or removal of<br>hairs or is not concerned | Increase in length, thickness or<br>density of hair at least on the<br>usual exposed areas of the<br>body [face (not limited to<br>beard/moustache area) | - | - | - |
| | enough about the overgrowth to use any form of hair removal | plus/minus arms] that requires<br>frequent shaving or use of<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial | | | |
| | | impact | | | |
| | zed by hair density or length beyon | | | | 1 |
| Hypohidrosis | - | Symptomatic; limiting instrumental ADL | Increase in body temperature;<br>limiting self care ADL | Heat stroke | Death |
| Definition: A disorder characteri | 1 | <u> </u> | | | 1 |
| Lipohypertrophy | Asymptomatic and covering <10% BSA | Covering 10 - 30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% BSA and associated tenderness and narcotics or NSAIDs indicated; lipohypertrophy; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by hypertrophy of the subcutan | eous adipose tissue at the site of | multiple subcutaneous injections of | of insulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by a change in the color of the | nail plate. | T | Т | |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the<br>nail bed from the nail plate or<br>nail loss; limiting instrumental<br>ADL | - | - | - |
| Definition: A disorder characteri | zed by loss of all or a portion of the | nail. | , | • | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by vertical or horizontal ridges | on the nails. | 1 | I | 1 |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensation | n in the skin. | T | Г | 1 |
| Palmar-plantar<br>erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling, blisters, bleeding, edema, or hyperkeratosis) with pain; limiting instrumental ADL | Severe skin changes (e.g., peeling, blisters, bleeding, edema, or hyperkeratosis) with pain; limiting self care ADL | - | - |
| | zed by redness, marked discomfort | | | reet. | |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by swelling due to an excessive | e accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Painless erythema and erythema covering <10% BSA | Tender erythema covering 10 - 30% BSA | Erythema covering >30% BSA and erythema with blistering; photosensitivity; oral corticosteroid therapy indicated; pain control indicated (e.g., narcotics or NSAIDs) | Life-threatening consequences; urgent intervention indicated | Death |

| | Sk | Skin and subcutaneous tissue disorders | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated;<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | - | - |
| Definition: A disorder character | ized by an intense itching sensation | | 1 | I | ' |
| Purpura | Combined area of lesions covering <10% BSA | Combined area of lesions covering 10 - 30% BSA; bleeding with trauma | Combined area of lesions covering >30% BSA; spontaneous bleeding | -<br>Dider lesions are usually a darker | -<br>ourple color |
| and eventually become a brown | | | | , | |
| Rash acneiform | Papules and/or pustules<br>covering <10% BSA, which may<br>or may not be associated with<br>symptoms of pruritus or<br>tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder character | ized by an eruption of papules and p | pustules, typically appearing in fac | ce, scalp, upper chest and back. | | |
| Rash maculo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering<br>>30% BSA with or without<br>associated symptoms; limiting<br>self care ADL | - | - |
| | ized by the presence of macules (fla | | nown as morbillform rash, it is one | of the most common cutaneous a | dverse |
| Scalp pain | upper trunk, spreading centripetally Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensation | n in the skin covering the top and | the back of the head. | Г | |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA; associated with ulceration | - | - |
| Definition: A disorder character | ized by the degeneration and thinning | ng of the epidermis and dermis. | T | T | |
| Skin hyperpigmentation | Hyperpigmentation covering <10% BSA; no psychosocial impact | Hyperpigmentation covering >10% BSA; associated psychosocial impact | - | - | - |
| Definition: A disorder character | ized by darkening of the skin due to | excessive melanin deposition. | | | |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | - | - | - |
| Definition: A disorder character | ized by loss of skin pigment. | | | | |
| Skin induration | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to slide skin, unable to pinch skin; limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| | ized by an area of hardness in the s | | T | T | |
| Skin ulceration | Combined area of ulcers <1 cm;<br>nonblanchable erythema of<br>intact skin with associated | Combined area of ulcers 1 - 2 cm; partial thickness skin loss involving skin or subcutaneous | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to or necrosis of | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or | Death |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | - | BSA with associated signs (e.g., 3) erythema, purpura, epidermal detachment and mucous el membrane detachment) m | | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment) | Death |
| Definition: A disorder characterize | ed by less than 10% total body ski | n area separation of dermis. The | syndrome is thought to be a hyper | sensitivity complex affecting the s | kin and the |
| mucous membranes. | | | _ | _ | |
| Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | - | - | - |
| Definition: A disorder characterize | ed by local dilatation of small vess | els resulting in red discoloration o | f the skin or mucous membranes. | | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characterize mucous membranes. | ed by greater than 30% total body | skin area separation of dermis. T | he syndrome is thought to be a hy | persensitivity complex affecting th | e skin and the |
| Urticaria | Urticarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 - 30% BSA; oral intervention indicated | Urticarial lesions covering >30%<br>BSA; IV intervention indicated | - | - |
| Definition: A disorder characterize | ed by an itchy skin eruption chara | cterized by wheals with pale interi | ors and well-defined red margins. | | |
| Skin and subcutaneous tissue disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Social circumstances | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 1 2 3 4 | | | |
| Menopause | Menopause occurring at age 46 - 53 years of age | Menopause occurring at age 40 - 45 years of age | Menopause occurring before age 40 years of age | - | - |
| Definition: A disorder characteriz | ed by the permanent cessation of | menses, usually defined by 12 co | nsecutive months of amenorrhea i | n a woman over 45 years of age. | |
| Social circumstances - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| procedures - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| 1 | | | disabling; limiting self care ADL | | |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by leakage of intravascular flui<br>ck syndromes, low-flow states, ische | · | • | • | |
| Flushing | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Symptomatic, associated with hypotension and/or tachycardia; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by episodic reddening of the fa | ice. | | | |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a localized collection of bloc | od, usually clotted, in an organ, sp | ace, or tissue, due to a break in th | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by an uncomfortable and temp | orary sensation of intense body w | armth, flushing, sometimes accom | panied by sweating upon cooling. | |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic<br>BP 140 - 159 mm Hg or<br>diastolic BP 90 - 99 mm Hg);<br>medical intervention indicated;<br>recurrent or persistent (>=24<br>hrs); symptomatic increase by<br>>20 mm Hg (diastolic) or to<br>>140/90 mm Hg if previously<br>WNL; monotherapy indicated | Stage 2 hypertension (systolic BP >=160 mm Hg or diastolic BP >=100 mm Hg); medical intervention indicated; more than one drug or more intensive therapy than previously used indicated Pediatric: Same as adult | Life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive crisis); urgent intervention indicated Pediatric: Same as adult | Death |
| Definition: A disorder characte | rized by a pathological increase in b | Pediatric: recurrent or persistent<br>(>=24 hrs) BP >ULN;<br>monotherapy indicated<br>lood pressure; a repeatedly eleval | | ng 140 over 90 mm Hg. | |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | 1 | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a blood pressure that is belo | ow the normal expected for an ind | ividual in a given environment. | | , |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by the loss of lymph fluid into t | | ĺ | | 1 |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery skin texture; papillary formation; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by excessive fluid collection in | tissues that causes swelling. | | | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | - | - |
| Definition: A disorder characte | rized by a cystic lesion containing ly | mph. | | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of ischemia managed non-<br>surgically and without permanent deficit | Recurring or prolonged (>=24<br>hrs) and/or invasive intervention<br>indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by impaired circulation to an ex | ktremity. | 1 | 1 | |
| Phlebitis | - | Present | - | - | - |
| Definition: A disorder characte | rized by inflammation of the wall of a | a vein. | | _ | |
| Superficial thrombophlebitis | - | Present | - | - | - |
| Definition: A disorder characte | rized by a blood clot and inflammation | on involving a superficial vein of th | e extremities. | | |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery) | Death |
| Definition: A disorder characteriz | ed by obstruction of the blood flow | in the superior vena cava. Signs | and symptoms include swelling ar | nd cyanosis of the face, neck, and | upper arms, |
| cough, orthopnea and headache | | | | T | |
| Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | Thrombosis (e.g., uncomplicated pulmonary embolism [venous], non-embolic cardiac mural [arterial] thrombus), medical intervention indicated | Life-threatening (e.g., pulmonary embolism, cerebrovascular event, arterial insufficiency); hemodynamic or neurologic instability; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream. | | |
| Vasculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the w | rall of a vessel. | | | |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of ischemia managed medically and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a decrease in blood supply | due to narrowing or blockage of a | visceral (mesenteric) artery. | | |
| Vascular disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |







NIH Publication No. 09-5410 Revised June 2010 Reprinted June 2010



## Appendix B: Pemphigus Disease Area Index

| - Skin | - Activity | - Damage | |
|---|---|---|---|
| Anatomical<br>Location | Erosion / Blisters or new erythema | | Post-inflammatory hyperpigmentation or |
| Location | • | Number | erythema from resolving lesion 0 absent |
| | 0 absent<br>1 1-3 lesions up to one > 2 cm in any diameter, none | lesions if 3 | 1 present |
| | > 6 cm | lesions II 3 | 1 present |
| | 2 2-3 lesions, at least two > 2 cm diameter, none > 6 | | |
| | cm | | |
| | 3 > 3 lesions, none > 6 cm diameter | | |
| | 5 > 3 lesions, and/or at least one > 6 cm | | |
| | 10 > 3 lesions, and/or at least one lesion > 16 cm | | |
| | diameter or entire area | | |
| Ears | | | |
| Nose | | | |
| Rest of the face | | | |
| Neck | | | |
| Chest | | | |
| Abdomen | | | |
| Back, buttocks | | | |
| Arms | | | |
| Hands | | | |
| Legs | | | |
| Feet | | | |
| Genitals | | | |
| Total skin | /120 | | /12 |
| - Scalp | | | |
| Scalp | Erosion/Blisters or new erythema | Number | Post-inflammatory hyperpigmentation or |
| F | • | lesions if 3 | erythema from resolving lesion |
| | 0 absent | | 0 absent |
| | 1 in one quadrant | | 1 present |
| | 2 two quadrants | | |
| | 3 three quadrants 4 affects whole skull | | |
| | 10 at least one lesion > 6 cm | | |
| Total Scalp (0-10) | /10 | | /1 |
| Mucous membran | | <u>l</u> | /1 |
| Anatomical | - | | |
| location | Erosion/Blisters | | |
| | 0 absent | Number | |
| | 1 1 lesion | lesions | |
| | 2 2-3 lesions | if 3 | |
| | 5 > 3 lesions or 2 lesions > 2 cm | | |
| | 10 entire area | | |
| Eyes | | | |
| Nose | | | |
| Buccal mucosa | | | |
| Hard palate | | | |
| Soft palate | | | |
| Upper gingiva | | | |
| Lower gingiva | | | |
| Tongue | | | |
| Floor of mouth | | | |
| Labial bucosa | | | |
| Posterior pharynx | | | |
| Anogenital | | | |
| Total Mucosa | /120 | | |

# Syntimmune, Inc.

### **CLINICAL STUDY PROTOCOL**

## A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

Medical Monitor: PPD

43 Thorndike Street, Cambridge, MA 01240

Phone: PPD extension PPD

Mobile: PPD

Original Protocol: 18 January 2017 Amendment 1.1: 21 March 2017

#### **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.
#### **SPONSOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the Investigator, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| PPU | |
|-----|--------------------------------|
| | March 21, 2017 |
| | Date of Signature (DD Mm YYYY) |

# PROCEDURES IN CASE OF EMERGENCY

#### Serious Adverse Events

Any death, serious adverse event (SAE)\* occurring in a subject while receiving study drug or within 7 days of receiving study drug, even though the event may not appear to be study drug related, must be promptly reported (within 24 hours) by telephone or electronic communication to the sponsor (or designee).

#### **Emergency Contact Information**



# **SAE CRITERIA**

- \* A <u>serious adverse event</u> (SAE) is any untoward medical occurrence that at any dose results in any of the following outcomes, regardless of relationship to study drug (see Section 11.3.1, Serious Adverse Events for additional information):
  - Death
  - Life-threatening adverse drug event
  - Inpatient hospitalization or prolongation of existing hospitalization
  - A persistent or significant disability/ incapacity
  - A congenital anomaly/birth defect
  - An important medical event that may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

Syntimmune, Inc.


Amendment 1.1 Final 21 March

# **INVESTIGATOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the sponsor, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonization Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

Nothing in this document is intended to limit the authority of a physician to provide emergency

| medical care under applicable regulations. | |
|---|---|
| Investigator Signature | Date of Signature<br>(DD Mm YYYY) |
| Name of Investigator (please print) | |

# 1 SYNOPSIS

| Study title | A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus) |
|---|---|
| Protocol number | SYNT001-103 |
| Number of study centers | Approximately 10 (US) |
| Clinical phase | Phase 1b |
| Study background | SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG immune complexes from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG containing immune complexes further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG immune complexes within and among compartments important in cellular immunity, it is further anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8+ and CD4+T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG and IC that are involved in many autoimmune conditions and dismantle their ability to cause disease. SYNT001 targets mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP). While current treatments for certain autoimmune disorders including chronic steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are frequently associated with significant adverse effects, an |

| | pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, leading to a significant decrease in total IgG, and thereby a corresponding decrease in the level of the pathogenic autoantibodies as well as the ICs to which they are associated, should lead to a decrease in the mucosal and cutaneous manifestations in subjects with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification. |
|---|---|
| Study rationale | This study is being conducted to further evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers. |
| Study objectives | Primary objective |
| | To evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus) |
| | Secondary objectives |
| | <ul> <li>To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels</li> <li>To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers: <ul> <li>Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM</li> <li>Albumin</li> </ul> </li> </ul> |
| | <ul> <li>Albumin</li> <li>To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers:</li> </ul> |
| | o Serum anti-desmoglein (Dsg) (1 and 3) antibody levels |
| | o Pemphigus Disease Area Index (PDAI) |
| | To assess immunogenicity (anti-SYNT001 antibodies) |
| | Exploratory objectives |
| | • To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including: |
| | <ul> <li>Serum anti-epithelial cell antibody (AECA) levels by indirect<br/>immunofluorescence</li> </ul> |
| | o Circulating immune complexes (CIC) |
| | o Complement component 3 (C3) |
| | <ul> <li>Exploratory biomarkers (FCGR2A (single nucleotide polymorphism-<br/>SNP), RNAseq, urine IgG)</li> </ul> |

# Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells SYNT001 levels in skin biopsies (optional)

- To characterize corticosteroid use during the study

#### Study design

Phase 1b, multicenter, open-label, safety, tolerability, and activity study

#### Methodology

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of subjects | Dose |
|--------|-----------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs, and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All safety data and any available and relevant PD data through Day 42 (2 weeks after the last subject's last dose in Cohort 1) will be reviewed by a dose escalation committee before Cohort 2 is initiated. Escalation to Cohort 2 will proceed if there are no concerning safety signals and the review of available and relevant PD data supports advancing to a higher dose. The dose for Cohort 2 will be finalized after review of the safety and PD data, but will not exceed 30 mg/kg. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule as Cohort 1.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33 and 56. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, and 42 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects also will return to the clinic on Day 56 (28 days after receiving their last dose of study drug) for an End-of-Study/Follow-Up visit.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, adverse event (AE) assessments, concomitant medication assessments, and electrocardiograms (ECG).

#### **Number of subjects**

Approximately 16; two cohorts of 8 subjects each. An additional cohort of up to 8 subjects may be enrolled. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects with pemphigus foliaceus may be enrolled.

# Diagnosis and main entry criteria

#### **Inclusion criteria:**

Subjects must meet the following criteria to be included:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq$  18 years of age at the time of screening;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal:
  - c. History of at least one positive tissue-based test (e.g., biopsy, direct immunofluorescence [DIF])
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose
     12 months prior to screening;

- b. If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
- c. If being treated with corticosteroids, must be  $\leq 1 \text{mg/kg/day}$  and stable (< 10% change in dose) for 2 weeks prior to screening;
- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 35.0 \text{ kg/m}^2$ ;
- 6. Has a negative urine pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through 60 days after the final study dose: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final study dose.

#### **Exclusion criteria:**

Subjects meeting any of the following criteria are to be excluded:

- 1. Subject unable or unwilling to comply with the protocol;
- Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG use within 60 days of screening;
- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;
- 8. Any exposure to an investigational drug or device within the 30 days prior to screening
- 9. Plasmapheresis or immunoadsorption within 60 days of screening

| | 10. Cellular therapy at any time prior to screening |
|---|---|
| | 11. Use of any immunosuppressive drugs apart from corticosteroids, |
| | azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of |
| | screening |
| | 12. Serum total IgG < 600 mg/dL; |
| | 13. Subject has any current medical condition that, in the opinion of the |
| | Investigator, may compromise their safety or compliance, preclude |
| | successful conduct of the study, or interfere with interpretation of the results |
| | (e.g., a significant pre-existing illness or other major comorbidity that the |
| | Investigator considers may confound the interpretation of the study results); |
| | 14. Any vaccination within 2 weeks of screening |
| Study drug, dosage, | SYNT001 |
| and administration | <b>Doses:</b> 10 mg/kg and 30 mg/kg. A third cohort of up to 8 subjects may be treated |
| | at another dose, with a maximum dose of 45 mg/kg, but may also be lower than |
| | 10 mg/kg or between 10 and 30 mg/kg, inclusive. |
| | SYNT001 is provided as a liquid at a nominal concentration of 50 mg/mL. |
| | SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for |
| | infusion. |
| | Route of administration: IV in 250 mL over 1 hour |
| Control, dose, and | Not applicable |
| route of | |
| administration | |
| <b>Duration of subject</b> | Up to 70 days (10 weeks): Screening of up to 2 weeks (14 days); dosing period |
| participation and | of 4 weeks (28 days); and 4 weeks (28 days) of follow-up |
| duration of study | |

# Prohibited

Concomitant

treatments

All treatments a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications may result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted.

Use of the following medications will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

#### Safety assessments

Safety assessments include AEs, serious adverse events (SAEs), PEs, vital sign measurements, clinical safety laboratory evaluations, ECGs, and reasons for treatment discontinuations due to toxicity. Safety assessments will be performed at specified time points and prior to discharge from the clinic. Vital sign measurements, including blood pressure, pulse rate, respiratory rate, and temperature will be monitored throughout the study. Pulse oximetry will be monitored during the study drug infusion and for 2 hours following the end of the infusion.

The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03) will be used for grading clinical and laboratory AEs.

| | The AE reporting period for a subject enrolled in the study begins when the subject provides informed consent and is continued for 28 days after the last dose of study drug. All AEs that occur in the enrolled subjects during the AE reporting period must be recorded, regardless of the relationship of the AE to study drug. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug should also be recorded. |
|---|---|
| Dose-escalation rules | Dose-limiting toxicity (DLT) will be defined generally as clinically significant, severe (Grade 3) AEs occurring in ≥ 2 subjects that are determined to be clinically significant and considered related to study drug. If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have |
| | Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and no further dose-escalation will occur. If the dose-escalation stopping rule is met in Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics data will be reviewed and a cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met after Cohort 1 (10 mg/kg), dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met in Cohort 2, all safety data and all available pharmacodynamics data will be reviewed and a cohort may be added at a dose at least 30% lower than the Cohort 2 dose. If the stopping rule is not met after Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data. |
| Study stopping rule | If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, any further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the next appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects. |
| Individual stopping rule | Dosing for any individual subject will be discontinued (i.e., further treatment with the study drug will not be given) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator and Medical Monitor, suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject may be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a |

| | significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus. |
|---|---|
| Pharmacokinetics | The PK of SYNT001 will be evaluated following the first and last (fifth) doses of SYNT001. |
| | Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. |
| | Study drug concentration will be used to calculate the following PK parameters: $t_{1/2},C_{max},T_{max},AUC_{0\text{-}24}$ , and $AUC_{0\text{-}\infty}$ . |
| Pharmacodynamics/<br>Activity | PD samples will be collected for analysis of IgG (serial assessment of IgG levels to identify C <sub>min</sub> , T <sub>min</sub> ); IgG1-4 subtype levels; IgA levels; IgM levels; albumin levels; anti-Dsg (1 and 3) antibody levels; serum AECA by direct immunofluorescence; CIC; C3; exploratory biomarkers ( <i>FCGR2A</i> SNP, RNAseq, urine IgG, CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T, monocytes, NK cells and B cells). |
| Immunogenicity | Up to 4 samples will be collected for immunogenicity analyses. Samples will be collected on Days 0 (pre-dose), 14, 28, and 56. |
| Skin biopsy | Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33 and 56 to analyze SYNT001 levels. |
| Photography | Photographs of active lesions will be taken at Day 0. Follow-up photographs of the same areas will be taken on Days 33 and 56. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. |
| Statistical methods | Sample size consideration |
| | Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives. |
| | Data presentations/Descriptive statistics |
| | Three populations will be employed in the analysis of study data. |
| | The intent-to-treat (ITT) population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population. |
| | The PK population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters. |

• The PD population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the PK and ITT populations, where appropriate.

#### Criteria for evaluation

| Objective | Endpoint |
|---|---|
| Primary | |
| Safety and tolerability of 5 once-<br>weekly IV infusions of SYNT001 to<br>subjects with pemphigus vulgaris or<br>foliaceus | AEs and clinical (safety) laboratory tests |
| Secondary | |
| PK of SYNT001 following a 1-hour IV infusion | $\begin{array}{ c c c c c }\hline PK \ parameters: t_{1/2}, C_{max}, T_{max}, \\ AUC_{0\text{-}24}, and \ AUC_{0\text{-}\infty}. \\ \end{array}$ |
| Effect of 5 once-weekly IV doses of SYNT001 on: • Total IgG (IgG1-4), IgA, IgM, and albumin • Serum anti-Dsg (1 and 3) antibodies | Changes in levels of IgG, IgG subtypes (IgG1-4), IgA, IgM, albumin, serum anti-Dsg (1 and 3) antibodies |
| Assess immunogenicity | Anti-SYNT001 antibodies |
| Disease Activity | PDAI Scores |
| Exploratory | |
| Effect of 5 once-weekly IV doses of SYNT001 on biomarkers including: • CIC • C3 • Serum anti-epithelial cell antibody (AECA) levels • Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG) • Immune phenotyping by flow cytometry | Changes in CIC; C3; AECA levels by indirect immunofluorescence; <i>FCGR2A</i> SNP; RNAseq; urine IgG, CD3+CD4+ T, CD3+CD8+ T, monocytes, NK cells and B cells; urine IgG levels; changes in blood transcriptome |
| Concomitant Treatment | Corticosteroid use during the study |
| SYNT001 levels in skin biopsies | Measures of SYNT001 levels in skin biopsies |

Treatment-emergent AEs (TEAEs) will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred

term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, or treatment discontinuation will be listed by subject, and cohort using SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken, and outcome.

Laboratory results will be summarized by time point and cohort. The incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the central laboratory. Vital sign measurements will be summarized by cohort at each scheduled time point using descriptive statistics.

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2},\,C_{max},\,T_{max},\,$  and area under the curve (AUC). PK parameters will be determined using non-compartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

PD results will be summarized by cohort. Descriptive statistics of PD parameters for SYNT001 will include mean, SD, CV, median, minimum, and maximum.

Immunogenicity results will be summarized by cohort. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

**Table 1:** Study Assessments

| Timepoint (Study Day) | Screen<br>-14 to -1 | 0 | 1<br>(±1<br>hr) | 2<br>(± 2<br>hr) | 5 <sup>p</sup> (±4 hr) | 7<br>(±4<br>hr) | 12 <sup>p</sup><br>(±6<br>hr) | 14<br>(±6<br>hr) | 19 <sup>p</sup><br>(±6<br>hr) | 21<br>(±6<br>hr) | 28<br>(±6<br>hr) | 29<br>(±1<br>hr) | 30<br>(±2<br>hr) | 33<br>(±4<br>hr) | 42<br>(±3<br>day) | Follow-Up<br>56<br>(±5 days) or<br>ET Visit | Extended<br>Follow-<br>up <sup>q</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | | | | | | | | | | |
| Demographics/Medical History | X | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | | | | | | |
| Physical Examination <sup>a</sup> | X | X | | | | X | | X | | X | X | | | | X | X | |
| Vital Signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Pulse Oximetry <sup>c</sup> | | X | | | | X | | X | | X | X | | | | | | |
| Clinical Safety Labs <sup>d</sup> | X | X | | | | X | | X | | X | X | | | X | X | X | |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | | | | | | | | X | |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | |
| 12-Lead ECG <sup>f</sup> | X | X | | | | | X | | | | X | | | | | X | |
| Tetanus & VZV antibodies <sup>g</sup> | | X | | | | | | | | | | | | | | X | X |
| PDAI Score | | X | | | | X | | X | | X | X | | | X | X | X | |
| PK Sampling <sup>h</sup> | | X | X | X | X | | | | | | X | X | X | X | | | |
| Immunogenicity <sup>i</sup> | | X | | | | | | X | | | X | | | | | X | |
| Study Drug Administration <sup>j</sup> | | X | | | | X | | X | | X | X | | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4) <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| CIC | | X | | | X | X | X | X | X | X | X | | | X | X | X | |
| Anti-Dsg (1 & 3) antibody titer | X | X | | | | X | | X | | | | | | X | | X | |
| C3 and AECA <sup>1</sup> | | X | | | | | | X | | | | | | X | | X | |
| FCGR2A <sup>m</sup> | | X | | | | | | | | | | | | | | | |
| RNAseq <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | |
| Urine IgG <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | |
| Immune phenotyping <sup>n</sup> | | X | | | | | | | | | X | | | | | | |
| Optional Skin Biopsy | | X | X | X | | | | X | | | | | | X | | X | |
| Photography <sup>o</sup> | | X | | | | | | | | | | | | X | | X | |
| Adverse Events | To be collected from the date that the ICF is signed until 28 days after last dose of study drug. | | | | | | | | | | | | | | | | |
| Concomitant Medications | | | To be | e collect | ted froi | n withi | in 14 de | avs prie | or to D | av 0 th | rough | 28 day | s after | last do | se of sti | ıdy drug. | |

Concomitant Medications

To be collected from within 14 days prior to Day 0 through 28 days after last dose of study drug.

ECG = electrocardiogram; ET= Early Termination; HIV = human immunodeficiency virus; ICF = informed consent form; PD = pharmacodynamic; PK = pharmacokinetic; VZV = varicella-zoster virus

Syntimmune, Inc.  Amendment 1.1 Final 21 March 2017


- a: Complete PE, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.
- b: **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. On Days 0, 7, 14, 21, and 28 vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- c: **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d: Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 6.7 for a complete list). Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42 and 56.
- e: **Pregnancy test:** To be performed at time of screening and prior to first dose of SYNT001 on Day 0 and on Day 56 (urine or serum test is acceptable, however, positive urine tests must be confirmed with serum testing.)
- f: Digital 12-lead ECG to be obtained after 5 minutes of rest in the supine position and in triplicate at least 1-2 minutes apart (see Section 6.6 for additional information). On Days 0 and 28 to be obtained 5 minutes after the completion of infusion. Day 12 ECG will be collected only if the visit is conducted at the study site.
- g: **Serology**: Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at 1 month after the Follow-Up visit (approximately 2 months after the subject's last dose); if still below the baseline value (or level of detection), the subject will be re-tested after another month (3 months after last dose). Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level on Day 56 and upon 2 retests (2 and 3 months following last dose of SYNT001), will be referred to their primary care physician for further management. See Section 6.7.3 for additional information.
- h: **PK:** Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. See Section 6.7.4 for additional information.
- i: Immunogenicity: Blood samples will be collected pre-dose when collected on dosing days. See Section 6.7.6 for additional information.
- j: Prior to **study drug infusion**, SYNT001 drug product is to be diluted in Dextrose 5% in Water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour using a 0.2-micron, inline filter. See Section 9 for additional information.
- k: Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, and IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 6.7.5 for additional information
- 1: Exploratory PD samples (C3 and AECA): collected pre-dose when collected on dosing days. See Section 6.7.5 for complete information.
- m: Samples to be collected and stored; pending review of clinical and pharmacodynamics assessments
- n: Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- o: Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 33 and 56. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- p: Visit Days 5, 12 and 19 may be conducted via at-home nursing in lieu of a subject visit to the study site.
- q: Extended follow-up visits will occur only if additional testing for anti-tetanus and/ or anti-VZV titers are required. These visits will occur as needed at approximately 2 months post last dose and 3 months post last dose.

Table 2: Timing Window Allowances for PK/PD Sampling, ECG, and Vital Sign Measurements

| Pharmacokinetic and Pharmacodynamic Sampling | |
|------------------------------------------------|-------------------------|
| Timepoint | Tolerance Window |
| 0 hour | −240 min to 0 hour |
| 5 minutes post end-of-infusion | ± 5 minutes |
| 2, 4, & 6 hours post end-of-infusion | ± 15 minutes |
| 24 hours post end-of-infusion | $\pm$ 60 minutes |
| 48 hours post end-of-infusion | ± 120 minutes |
| ECG | |
| Timepoint | <b>Tolerance Window</b> |
| 5 minutes post end-of-infusion | ± 10 minutes |
| Vital Signs <sup>a</sup> | |
| Timepoint | <b>Tolerance Window</b> |
| 0 hour | −240 min to 0 hour |
| 15, 30, and 45 minutes after start of infusion | ± 5 minutes |
| 60 minutes after start of infusion | ± 10 minutes |
| 30, 60 and 120 minutes post end-of-infusion | ± 10 minutes |

a: Vital signs to include blood pressure, pulse rate, respiratory rate, oral temperature, and pulse oximetry.

# TABLE OF CONTENTS

| PROCE | EDURES IN CASE OF EMERGENCY | 3 |
|--------|---------------------------------------------|----|
| INVES' | TIGATOR SIGNATURE | 4 |
| 1 S | YNOPSIS | 5 |
| LIST O | OF ABBREVIATIONS | 24 |
| 2 B | ACKGROUND AND RATIONALE | 26 |
| 2.1 | Study Rationale | 27 |
| 2.2 | Selection of Doses in this Study | |
| 2.3 | Compliance Statement | |
| 3 ST | TUDY OBJECTIVES | 29 |
| 3.1 | Primary Objective | 29 |
| 3.2 | Secondary Objectives | 29 |
| 3.3 | Exploratory Objectives | 29 |
| 4 ST | TUDY DESIGN | 30 |
| 4.1 | Study Sites | 30 |
| 4.2 | Study Endpoints | 30 |
| 4.3 | Overview of Study Design | 31 |
| 4.4 | Randomization and Blinding | 33 |
| 5 ST | TUDY POPULATION | 34 |
| 5.1 | Target Population | 34 |
| 5.2 | Inclusion Criteria | 34 |
| 5.3 | Exclusion Criteria | 35 |
| 6 ST | TUDY PROCEDURES | 37 |
| 6.1 | Informed Consent | 37 |
| 6.2 | Demographics and Medical History | 37 |
| 6.3 | Physical Examination. | |
| 6.4 | Pemphigus Disease Area Index (PDAI) Scoring | 37 |
| 6.5 | Vital Sign Measurements | |
| 6.6 | | |
| 6.7 | • | |
| | 6.7.1 Pregnancy Testing | |
| | 6.7.2 Virology | 40 |

| | | 6.7.3 | Serum Tetanus Antibody and Varicella-Zoster Virus Antibo | dy Testing40 |
|---|---|---|---|---|
| | | 6.7.4 | Pharmacokinetics (PK) Sampling | 41 |
| | | 6.7.5 | Pharmacodynamic Sampling | 41 |
| | | 6.7.6 | Immunogenicity Testing | 42 |
| | 6.8 | Study | y Drug Administration | 43 |
| | 6.9 | Prior | and Concomitant Medications | 43 |
| | 6.10 | Adve | erse Event Assessments | 43 |
| | 6.11 | Photo | ographs | 44 |
| | 6.12 | Skin | Biopsy | 44 |
| 7 | STUDY ASSESSMENTS45 | | | |
| | 7.1 | Scree | ening Period: Day -14 to Day -1 | 45 |
| | 7.2 | | Ilment and First Treatment: Day 0 | |
| | 7.3 | Follo | w-up: Day 1 | 47 |
| | 7.4 | Follo | w-up: Day 2 | 47 |
| | 7.5 | Follo | w-up: Day 5 | 48 |
| | 7.6 | Treat | ment Day 7 (Dose 2) | 48 |
| | 7.7 | Dose | 2 Follow-up Day 12 | 49 |
| | 7.8 | Treat | ment Day 14 (Dose 3) | 49 |
| | 7.9 | Dose | 3 Follow-up Day 19 | 51 |
| | 7.10 | Treat | ment Day 21 (Dose 4) | 51 |
| | 7.11 | Treat | ment Day 28 (Dose 5) | 52 |
| | 7.12 | Follo | w-up Day 29 | 53 |
| | 7.13 | Follo | w-up Day 30 | 54 |
| | 7.14 | 4 Follow-up Day 33 | | |
| | 7.15 | Follo | w-up Day 42 | 55 |
| | 7.16 | Follo | w-up Day 56 (End-of-Study) or Early Termination Visit | 55 |
| | 7.17 | Exte | nded Follow-up Visits | 56 |
| 8 | REMOVING SUBJECTS FROM STUDY57 | | | |
| | 8.1 | Subje | ect Withdrawal | 57 |
| | 8.2 | Study | y Discontinuation | 58 |
| | 8.3 | Repla | acements | 58 |
| | 8.4 | Stopp | ping Rule | 58 |
| | | 8.4.1 | Dose-Escalation Stopping Rule | 58 |
| | | 8.4.2 | Study Stopping Rule | 59 |
| | | 8.4.3 | Individual Stopping Rule | 59 |
| 9 | ST | UDY D | RUG | 60 |
| | 9.1 | SYN | T001 | 60 |

| | 9.2 | Cohort | Dosing | 60 |
|---|---|---|---|---|
| | 9.3 | | g of Dosing | |
| | 9.4 | Identit | y of Investigational Products | 60 |
| | 9.5 | Investi | gational Product Retention at Study Site | 61 |
| | 9.6 | Warnii | ngs and Precautions | 61 |
| | | 9.6.1 | Infusion Reaction | 61 |
| | | 9.6.2 | Potential Immune Effects | 66 |
| 0 | CC | NCOMI' | FANT MEDICATION AND TREATMENT | 67 |
| 1 | SA | FETY | | 69 |
| | 11.1 | Safety | Parameters | 69 |
| | 11.2 | Advers | se Event Definition | 69 |
| | 11.3 | Evalua | ting Adverse Events | 70 |
| | | 11.3.1 | Serious Adverse Events | 70 |
| | | 11.3.2 | Overdose | 71 |
| | | 11.3.3 | Non-Serious Adverse Events | 71 |
| | | 11.3.4 | Protocol-Related Adverse Events | 71 |
| | | 11.3.5 | Assessment of Causality | 71 |
| | | 11.3.6 | Recording Adverse Events | 72 |
| | | 11.3.7 | Planned Hospitalization | 72 |
| | | 11.3.8 | Reporting Pregnancies | 73 |
| | | 11.3.9 | Serious Adverse Event Reporting | 73 |
| | | 11.3.9.1 | Governing Regulatory Requirements | 73 |
| | | 11.3.9.2 | Time Frame for Reporting | 74 |
| | | 11.3.9.3 | Information to be Provided by the Investigator | 75 |
| | | | Regulatory Reporting | |
| | | 11.3.11 | Follow-up Information on a Serious Adverse Event (SAE) | 77 |
| | 11.4 | Other S | Safety Considerations | 77 |
| | | 11.4.1 | Laboratory Data | 77 |
| | | 11.4.2 | Medication Errors | 77 |
| | | 11.4.3 | Follow-Up of Adverse Events | 77 |
| | 11.5 | Safety | Monitoring for Dose Escalation | 78 |
| 12 | ST | ATISTIC | AL CONSIDERATIONS | 79 |
| | 12.1 | Genera | ıl Design | 79 |
| | 12.2 | Sample | e Size Justification | 79 |
| | 12.3 | Statisti | cal Considerations | 79 |
| | | 12.3.1 | Study Populations | 79 |
| | | 12.3.2 | Subject Accountability, Demographics, and Baseline Characteristic | cs 80 |

| | | 12.3.3 | Concomitant Medications | 80 |
|----|------|---------|----------------------------------------------|-------|
| | 12.4 | Planne | ed PK Analysis | 80 |
| | 12.5 | Safety | Data | 81 |
| | 12.6 | Pharm | acodynamic/Activity Data | 81 |
| | 12.7 | Immu | nogenicity Data | 81 |
| | 12.8 | Interin | n Analysis | 82 |
| 13 | DA | TA QUA | ALITY ASSURANCE | 83 |
| 14 | ST | UDY AD | MINISTRATION | 84 |
| | 14.1 | Study | Administrative Structure | 84 |
| | 14.2 | Ethica | l Conduct of the Study | 84 |
| | 14.3 | Inform | ned Consent (ICF) | 84 |
| | 14.4 | Institu | tional Review Board | 85 |
| | 14.5 | Dose I | Escalation Committee | 85 |
| | 14.6 | Future | Use of Subject Samples | 86 |
| 15 | CC | NDITIO | NS FOR MODIFYING THE PROTOCOL | 87 |
| 16 | CC | NDITIO | NS FOR TERMINATING THE STUDY | 88 |
| 17 | ST | UDY DC | CUMENTATION, CRFS, AND RECORD KEEPING | 89 |
| | 17.1 | Investi | gator's Files and Retention of Documents | 89 |
| | 17.2 | Source | Documents and Background Data | 89 |
| | 17.3 | Audits | and Inspections | 90 |
| | 17.4 | Electro | onic Case Report Forms | 91 |
| 18 | MO | ONITOR | ING THE STUDY | 92 |
| 19 | CC | NFIDEN | ITIALITY OF TRIAL DOCUMENTS AND SUBJECT RECO | RDS93 |
| 20 | PU | BLICAT | ION OF DATA AND PROTECTION OF TRADE SECRETS | 94 |
| 21 | RF | FERENC | TES | 95 |

| Table 1: | Study Assessments | 16 |
|---|---|---|
| Table 2: | Timing Window Allowances for PK/PD Sampling, ECG, and Vital Sign | |
| | Measurements | 18 |
| Table 3: | Clinical Laboratory Panels | 39 |
| Table 4: | Pharmacodynamic/ Activity Assessments | 42 |
| Table 5: | Grading and Management of Allergic or Infusion-Related Reactions | 65 |
| Table 6: | Study Administrative Structure | |
| • | Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions Management of Severe (Grade 3 or higher) Infusion Reactions | |
| LIST OF A | APPENDICES | |
| Appendix A | A: NCI CTCAE, Version 4.03 | 96 |
| Appendix E | 3: Pemphigus Disease Area Index | 97 |

#### LIST OF ABBREVIATIONS

ADA Anti-drug antibodies

AE Adverse event

AECA Anti-epithelial cell antibody
ALT Alanine aminotransferase
ANA Antinuclear antibody
AST Aspartate aminotransferase
ATC Anatomical therapeutic chemical

 $AUC_{0-24}$  Area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose

 $AUC_{0-\infty}$  Area under the plasma concentration-time curve from pre-dose (time 0) to infinity

BLQ Below the limit of quantification

BMI Body mass index
BUN Blood urea nitrogen

CAR-T Chimeric antigen receptor and T-cell

CFR Code of Federal Regulations
C3 Complement component 3
CBC Complete blood count

CIC Circulating immune complexes

CIDP Chronic inflammatory demyelinating polyneuropathy

C<sub>max</sub> Maximum plasma concentration determined directly from the concentration-time profile

CRO Contract research organization

CV Coefficient of variation

CVID Common variable immune deficiency

DEC Dose escalation committee
D5W Dextrose 5% in Water
DIF Direct immunofluorescence
DNA Deoxyribonucleic acid
ECG Electrocardiogram

eCRF Electronic case report form
ESR Erythrocyte sedimentation rate
FcGR2a Fc Gamma R2a receptor
FcRn Neonatal Fc receptor

FDA Food and Drug Administration

GCP Good Clinical Practice

GI Gastrointestinal
HBV Hepatitis B virus
HCV Hepatitis C virus

HIPAA Health Insurance Portability and Accountability Act

HIV Human immunodeficiency virus

IB Investigator's brochure IC Immune complex

ICF Informed consent form

ICH International Conference on Harmonization

IgA Immunoglobulin A
IgG Immunoglobulin G
IgG1-4 Immunoglobulin G1-G4
IgM Immunoglobulin M
IL-12 Interleukin 12

IND Investigational new drug
IRB Institutional review board

ITT Intent-to-treat
IUD Intrauterine devices

IV Intravenous

IVIG Intravenous immunoglobulin

MedDRA Medical Dictionary for Regulatory Activities

NHL Non-Hodgkin lymphoma
PD Pharmacodynamics
PE Physical examination
PK Pharmacokinetic
RBC Red blood cells
RNAseq RNA sequencing

QTcF Corrected QT interval using Fridericia's formula

SAE Serious adverse event SAP Statistical analysis plan SAS Statistical Analysis System

SD Standard deviation

SNP Single nucleotide polymorphism

SOC System Organ Class

SOP Standard operating procedures

SYNT001 A humanized, affinity matured IgG4-kappa monoclonal antibody

 $t_{1/2}$  Half-life

TEAE Treatment-emergent adverse event

T<sub>max</sub> Observed time to reach peak plasma concentration

TNF Tumor necrosis factor ULN Upper limit of normal

UNS Unscheduled

VZV Varicella-zoster virus

WAIHA Warm antibody autoimmune hemolytic anemia

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

#### 2 BACKGROUND AND RATIONALE

SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG ICs from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG-containing ICs further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen-presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG ICs within and among compartments important in cellular immunity, it is anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8<sup>+</sup> and CD4<sup>+</sup> T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG that are involved in certain autoimmune conditions and dismantle their ability to cause disease.

SYNT001 targets key mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP).

While current treatments for certain autoimmune disorders, including high-dose steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are associated with significant adverse effects, as well as delayed or non-durable responses.

Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies have been shown to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, which significantly decreases total IgG, including a corresponding decrease in the level of the pathogenic autoantibodies and the ICs to which they are associated, may lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification.

# 2.1 Study Rationale

This study is being conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers.

# 2.2 Selection of Doses in this Study

The planned dose levels of SYNT001 for this Phase 1b safety and proof-of-concept study of 10 mg/kg and 30 mg/kg were selected from careful review of the safety, tolerability, and PD effect on total IgG levels after single and repeat dosing of SYNT001 in non-human primates (NHPs), as well as the safety, tolerability, and PD effect on total IgG levels after single ascending doses of SYNT001 in healthy volunteers. In addition, further consideration was given to the desired level of FcRn blockade to achieve suppression of IgG to a range that has been previously correlated with disease remission. Further, we considered the potential effects of inhibiting FcRn function as they relate to immune complex associated innate and adaptive immunity in choosing these dose levels based upon exploratory studies of a single ascending dose of SYNT001 in healthy volunteers. From the NHP studies, single doses of SYNT001 produced a dose-dependent decrease in total IgG and a further decrease was seen with repeated weekly doses up to a maximum 70% reduction at 100 mg/kg. This magnitude of total IgG reduction is approaching the expected maximal effect of 100% inhibition of FcRn function based on murine studies also performed by Syntimmune and others [Roopenian 2003, Nixon 2015]. In the recently completed Phase 1a trial with SYNT001 in healthy volunteers a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the NHP studies further reductions are expected following multiple dosing. A comparable decrease in pathogenic autoantibodies is also anticipated.

In the NHP studies, relevant adverse effects, mild-to-moderate infusion reactions, were observed only after the third weekly IV administration, concurrent with the development of anti-SYNT001 antibodies. In the recently completed Phase 1a healthy male volunteer study, the doses of SYNT001 up to and including 30 mg/kg have been well tolerated. There were no dose limiting toxicities, serious adverse events, or any other safety concerns identified. No AEs were observed in the 1 and 3 mg/kg dose cohorts. A single Grade 2 AE was observed; a headache in the 10 mg/kg cohort, treated with acetaminophen. Other subjects had mild (Grade 1) AEs at 10 mg/kg. In Cohort 4 (30 mg/kg), 5 subjects received SYNT001. All five subjects experienced AEs; all were mild (Grade 1), transient and resolved spontaneously without intervention. Therefore, it is anticipated that the doses selected for this study should be well tolerated and have clinically relevant PD effects in patients with chronic pemphigus (vulgaris or foliaceus). For a summary of

findings from the single dose, clinical study in healthy subjects and further details on the nonclinical findings, please refer to the SYNT001 Investigator's Brochure.

# 2.3 Compliance Statement

This study will be conducted in compliance with Good Clinical Practice (GCP), including the International Conference on Harmonisation (ICH) Guidelines and FDA regulations, consistent with the principles outlined in the Declaration of Helsinki. In addition, the Investigator agrees to adhere to all applicable local laws and regulatory requirements relevant to the use of new therapeutic agents.

The study will be conducted in compliance with the protocol. The appropriate Institutional Review Boards (IRBs) must approve the protocol, any amendments, and the subject informed consent form (ICF) prior to implementation.

Freely given written informed consent must be obtained from every subject prior to participation in this clinical trial. As part of this procedure, the Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or AEs that may occur. The study subject should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The Investigator or designee will provide the Sponsor with a copy of the IRB-approved informed consent form prior to the start of the study. The rights, safety, and well-being of participating subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (e.g., loss of medical licensure, debarment).

#### 3 STUDY OBJECTIVES

# 3.1 Primary Objective

The primary objective of this study is to evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus).

# 3.2 Secondary Objectives

The secondary objectives of this study are as follow:

- To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers:
  - o Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM
  - o Albumin
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers:
  - o Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
  - o Pemphigus Disease Area Index (PDAI)
- To assess immunogenicity (anti-SYNT001 antibodies)

#### 3.3 Exploratory Objectives

The exploratory objectives of this study are as follow:

- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including:
  - o Serum anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence
  - o Circulating immune complexes (CIC)
  - o Complement component 3 (C3)
  - Exploratory biomarkers (FCGR2A single nucleotide polymorphism-SNP, RNAseq, urine IgG)
  - Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
  - o SYNT001 levels in skin biopsies (optional)
- To characterize corticosteroid use during the study

#### 4 STUDY DESIGN

# 4.1 Study Sites

This study will be conducted at approximately 10 sites in the United States (US).

#### 4.2 Study Endpoints

**Primary Outcome Measures:** Assessment of safety data (adverse events [AEs], serious adverse events [SAEs], vital sign measurements, ECGs and clinical laboratory tests) will be the primary safety measure.

#### **Secondary Outcome Measures**

#### Pharmacokinetics:

Half-life (t<sub>1/2</sub>), maximum plasma concentration determined directly from the concentration-time profile (C<sub>max</sub>), observed time to reach peak plasma concentration (T<sub>max</sub>), area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose (AUC<sub>0-24</sub>), and area under the plasma concentration-time curve from pre-dose (time 0) to infinity (AUC<sub>0-∞</sub>)

#### PD Biomarkers:

- Ig Assessments: Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o IgA levels
  - o IgM levels
- Albumin levels

#### Disease activity markers:

- Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
- Pemphigus Disease Area Index (PDAI) scores

#### Immunogenicity:

• Anti-SYNT001 antibodies

#### **Exploratory Outcome Measures**

Biomarkers, including:

- CIC
- C3
- Serum AECA levels
- Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG)

- Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- SYNT001 levels in skin biopsies (optional)

#### **Concomitant Treatments**

Corticosteroid use

Further details on the statistical and analytical plan for these endpoints are available in Section 12, Statistical Considerations.

# 4.3 Overview of Study Design

This will be a multicenter, open-label study to assess the safety, tolerability, activity, PK, PD, and immunogenicity of 5 once-weekly IV infusions of SYNT001 to subjects with chronic pemphigus (vulgaris or foliaceus).

Planned doses of SYNT001 to be studied are 10 mg/kg and up to 30 mg/kg. Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 10 mg/kg or up to 30 mg/kg. Based on review of safety, PD, and clinical outcomes of the first cohort, the dose for the second cohort may be adjusted, but with a maximum dose of 30 mg/kg. Based on review of safety, PD and clinical outcomes from these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of<br>Subjects | Dose |
|--------|--------------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All data through Day 42

(2 weeks after the last subject's last dose in Cohort 1) will be reviewed before Cohort 2 is initiated. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule.

Safety evaluations will be conducted by a dose escalation committee (DEC). The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions. Dosing and dose escalation will proceed if the DEC has determined that it would be safe and appropriate to do so. In addition, over the course of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33 and 56. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, and 42 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects also will return to the clinic on Day 56 (28 days after receiving their last dose of study drug) for an End-of-Study/Follow-Up visit.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, AE assessments, concomitant medication assessments, and electrocardiograms (ECG).

**Note**: No vaccinations may be given from within 2 weeks of screening until 2 months following the last dose of study drug.

# 4.4 Randomization and Blinding

This is an open-label study.

#### 5 STUDY POPULATION

# 5.1 Target Population

This study will be conducted in approximately 16 male and female subjects (2 cohorts of 8 subjects each) with a confirmed diagnosis of pemphigus (vulgaris or foliaceus); however, a third cohort of up to 8 subjects may be added. Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through 28 days after their last dose. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects may be enrolled with pemphigus foliaceus.

#### 5.2 Inclusion Criteria

A subject must meet the following criteria to be eligible for the study:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq$  18 years of age;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal;
  - c. History of at least one positive tissue based test (biopsy, DIF)
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose > 12 months prior to screening;
  - If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
  - c. If being treated with corticosteroids, must be ≤ 1mg/kg/day and stable (< 10% change in dose) for 2 weeks prior to screening;

- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 35.0 \text{ kg/m}^2$ ;
- 6. Has a negative urine pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through 60 days after the final study dose: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final study dose.

# 5.3 Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

- 1. Unable or unwilling to comply with the protocol;
- Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG treatment within 60 days of screening;

- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;
- 8. Any exposure to an investigational drug or device within 30 days prior to screening;
- 9. Plasmapheresis or immunoadsorption within 60 days of screening
- 10. Cellular therapy at any time prior to screening
- 11. Use of any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of screening;
- 12. Serum total IgG < 600 mg/dL;
- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (e.g., a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results);
- 14. Any vaccination within 2 weeks of screening

#### 6 STUDY PROCEDURES

#### 6.1 Informed Consent

All subjects must take part in the informed consent process. Adequate time must be allowed for the subject to ask questions and make a voluntary decision. No protocol-specific procedures, including screening procedures, are to be performed until the subject has signed and dated an IRB-approved ICF. Subjects may withdraw consent at any time. Participation in the study may be terminated at any time without the subject's consent as determined by the Investigator.

# 6.2 Demographics and Medical History

Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and eCRF. Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery and concomitant treatments.

# 6.3 Physical Examination

A complete physical examination will be performed as outlined in Table 1. The complete PE will include measurements of weight (in kg) and height (in cm; height to be measured only at screening visit) and a review of the following body systems:

- General appearance
- Head, eyes, ears, nose, and throat
- Neck
- Respiratory
- Cardiovascular
- Abdomen
- Neurologic
- Extremities
- Dermatologic
- Lymphatic

Any abnormal and clinically significant findings from the PE must be recorded in the appropriate eCRF. Findings at screening and Day 0 (pre-dose) will be recorded as medical history.

# 6.4 Pemphigus Disease Area Index (PDAI) Scoring

Pemphigus severity and disease activity will be measured using the PDAI. See Appendix B.

# 6.5 Vital Sign Measurements

Vital sign measurements will be collected after the subject has been sitting for 5 minutes. Vital sign assessments will include measurements of sitting blood pressure (mm Hg), heart rate (beats
per minute), respiration rate (breaths per minute), oral temperature (Celsius). Abnormal results are to be repeated after 5 minutes of rest. Pulse oximetry (%) also is to be measured. See Table 2 for timing window allowances with respect to measurement collection.

On Days 0, 7, 14, 21, and 28, vital sign measurements are to be obtained immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion. Details on the management of mild to moderate and severe infusion reactions can be found in Figure 1 and Figure 2. Abnormalities in vital sign measurements will be graded in severity per the NCI CTCAE scale Version 4.03.

Subjects should be seated quietly for at least 5 minutes in a chair with their backs supported, their feet flat on floor (legs uncrossed), and their arms bared on a hard surface, with the arm slightly abducted and bent, with palm up and the midpoint of upper arm at heart level. Correct cuff and bladder size should be utilized and the same cuff and arm should be used per subject throughout study.

#### 6.6 12-Lead Electrocardiogram (ECG)

Digital 12-lead ECG measurements will be obtained at screening, on Days 0 and 28 at 5 minutes after the completion of the infusion and at the Day 56 (Follow-Up) Visit. Subjects who conduct their Day 12 visit at the investigative site, as opposed to an at-home nurse visit, will have an additional ECG performed. ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each 1 to 2 minutes apart. See Table 2 for timing window allowances with respect to performing ECG.

The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant.

Normal QTcF is  $\leq 450$  msec.

Abnormalities in the ECG that appear following therapy or that result in clinical signs and symptoms are considered clinically significant for the purposes of this study and will be recorded on the AE eCRF.

#### 6.7 Clinical Laboratory Measurements

Collection time for all safety, PD, and exploratory labs are outlined in Table 1.

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and anti-drug antibody samples) will be performed using established methods by a central laboratory. Safety laboratory panels are defined as listed in Table 3. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and anti-drug antibody samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42 and 56. The total blood draw for each subject who completes the study at Day 56, will be approximately 311 mL. Please refer to the Laboratory Manual for more information.

**Table 3:** Clinical Laboratory Panels

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| CBC with differential Erythrocyte Sedimentation Rate (ESR) | <ul> <li>Albumin</li> <li>Alkaline phosphatase</li> <li>ALT</li> <li>AST</li> <li>BUN</li> <li>Calcium</li> <li>Carbon dioxide</li> <li>Chloride</li> <li>Creatinine</li> <li>Glucose</li> <li>LDH</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total and direct bilirubin</li> <li>Total protein</li> <li>Uric acid</li> <li>C-Reactive Protein</li> </ul> | <ul> <li>Appearance</li> <li>Color</li> <li>pH</li> <li>Specific gravity</li> <li>Ketones</li> <li>Protein</li> <li>Glucose</li> <li>Nitrite</li> <li>Urobilinogen</li> <li>Blood/hemoglobin</li> <li>Leukocyte esterase</li> <li>Bilirubin</li> <li>Microscopic examination of sediment: only if the results of the urinalysis dipstick evaluation are positive for blood/hemoglobin</li> </ul> |
| Virology | | |
| <ul><li>Hepatitis C</li><li>Hepatitis B</li></ul> | | |

- HIV
- VZV
- Tetanus

ALT = alanine aminotransferase; AST = aspartate aminotransferase; CBC = complete blood count; BUN = blood urea nitrogen; HIV = human immunodeficiency virus; LDH = lactate dehydrogenase; VZV = varicella-zoster virus

Abnormalities in clinical laboratory tests that are considered clinically significant are to be recorded on the AE electronic case report form (eCRF) page. Laboratory results will be graded using the NCI CTCAE, Version 4.03. If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as an SAE (see Section 11.3.1).

#### 6.7.1 Pregnancy Testing

Pregnancy testing will be performed for women of childbearing potential at screening and prior to first dose of SYNT001 on Day 0 and Day 56 (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing.)

#### 6.7.2 Virology

Testing for HCV antibody, hepatitis B surface antigen, and HIV antibody will be performed at screening.

#### 6.7.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

Samples for serum tetanus antibody and varicella-zoster virus antibody testing are to be collected at baseline (pre-dose, Day 0) and on Day 56 (Follow-Up visit). Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. Specifically, if the baseline VZV titer is above the detectable level, but tetanus is not, only the VZV antibody titer will be tested on Day 56. If the Day 56 results are below the baseline value, defined as greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at 1 month after the Follow-Up visit (approximately 2 months after the subject's last dose); if still below the baseline value (or level of detection), the subject will be re-tested after another month (3 months after last dose). Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level on Day 56 and upon 2 retests (2 and 3 months following last dose of SYNT001), will be referred to their primary care physician for further management.

#### 6.7.4 Pharmacokinetics (PK) Sampling

Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. The actual time and date of each blood draw is to be recorded.

Study drug concentration will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-24}$ , and  $AUC_{0-\infty}$ .

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual

#### 6.7.5 Pharmacodynamic Sampling

PD samples will be collected for analyses throughout the study. On Days 0, 7, 14, 21, and 28, samples should be collected prior to infusion of study drug. Measurements for albumin PD biomarkers will be derived from the clinical safety laboratory results. Samples for each type of PD will be collected according to the schedule shown in Table 4.

Table 4: Pharmacodynamic/ Activity Assessments

| Parameter | Collection Timepoints |
|---|---|
| IgG, IgG subtypes (IgG1-4), IgA, IgM | Screening, and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, and 56 |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, and 56 |
| Albumin | Screening, and Days 0, 7, 14,21, 28, 33, 42, and 56 |
| Anti-Dsg (1 and 3) antibody titer | Screening, Days 0, 7, 14, 33, and 56 |
| <ul> <li>Complement component 3 (C3)</li> <li>Anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence</li> </ul> | Days 0, 14, 33, and 56 |
| Exploratory biomarker (RNAseq, Urine IgG) | Days 0, 14, 33, and 56 |
| Immune phenotyping by flow cytometry for<br>measurement of CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T,<br>monocytes, NK cells and B cells | Days 0 and 28 |
| Exploratory biomarker (FCGR2A SNP) | Day 0 |

See Table 2 for timing window allowances with respect to measurement collection. Detailed instructions for sample collection (including collection tubes) and preparation will be provided in a separate laboratory manual.

#### 6.7.6 Immunogenicity Testing

Up to 4 serum samples will be collected for immunogenicity analyses. Samples will be collected on Days 0 (pre-dose), 14, 28, and 56.

SYNT001 is being developed for the acute and chronic therapy of autoimmune disorders. Although SYNT001 is a humanized IgG4 monoclonal antibody, exposure to SYNT001 in clinical trials could result in the development of anti-drug antibodies (ADAs), with potential consequences ranging from neutralization or lessening of drug efficacy to safety consequences such as allergic reactions. Testing will first detect binding ADAs, then, for all confirmed positive samples, there will be testing for neutralizing effects.

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

#### 6.8 Study Drug Administration

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute IV infusions of SYNT001 10 mg/kg or up to 30 mg/kg. SYNT001 will be given as a 250-mL IV infusion over 1 hour using a 0.2-micron, inline filter. Based on review of safety data, as well as available and relevant PD results, and clinical outcomes of Cohort 1, a decision about proceeding with Cohort 2 will be made. Based on review of all safety data, available PD results, and clinical outcomes of these 2 cohorts, a third cohort of 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort No. | Study Drug | Dose Level (mg/kg/dose) |
|------------|------------|-------------------------|
| 1 | SYNT001 | 10 mg/kg |
| 2 | SYNT001 | 30 mg/kg |

See Section 9.1 for dosing schedule.

#### 6.9 Prior and Concomitant Medications

All medications a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented on the source document and eCRF.

Note: No vaccinations may be given from within 2 weeks of screening until 2 months following the last dose of study drug.

#### 6.10 Adverse Event Assessments

Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form throughout their participation in the study, including a period of 28 days after study drug dosing. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE.

Clinical AEs will be graded using the NCI CTCAE, Version 4.03 (Appendix A).

**Note**: AEs resulting in a subject's permanent discontinuation from the study, regardless of seriousness or relationship to study drug, MUST be promptly reported to the sponsor. Additionally, subjects must be followed until return to normal and/or resolution of the AE.

See Section 11 for more information.

#### 6.11 Photographs

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33 and 56. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

### 6.12 Skin Biopsy

Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33 and 56 to analyze SYNT001 levels.

#### 7 STUDY ASSESSMENTS

#### 7.1 Screening Period: Day -14 to Day -1

Informed consent must be obtained before any study-specific samples are taken or study-specific tests or evaluations are conducted. The following assessments at the screening visit are to occur within 14 days before dosing. Study eligibility will be based on satisfying all the study inclusion and exclusion criteria.

At the screening visit, information will be collected and subjects will have clinical evaluations as follows:

- Informed consent (Section 6.1)
- Medical history and demographic data (Section 6.2)
- Review inclusion and exclusion criteria (Section 5.2, Section 5.3)
- Complete PE, including height and weight (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Section 6.6)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Hepatitis and HIV screen (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.2 Enrollment and First Treatment: Day 0

Study Day 0 is defined as the date the subject is administered their first dose of study drug. On Day 0, subjects will be asked to come to the clinic and the following procedures will be performed prior to the first dose of study drug:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)

- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody (Section 6.7)
- PDAI Score (Section 6.4)
- PK baseline sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - FCGR2A SNP
  - RNAseq
  - Urine IgG
  - Immune phenotyping
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral

temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)

- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.3 Follow-up: Day 1

On Day 1 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.4 Follow-up: Day 2

On Day 2 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.5 Follow-up: Day 5

On Day 5 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 0), subjects may return to the clinic or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.6 Treatment Day 7 (Dose 2)

On Day 7 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion

and at completion of the infusion (Section 6.5)

- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.7 Dose 2 Follow-up Day 12

On Day 12 ( $\pm$  6 hours) the subject may will return to the clinic, or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- If visit performed at the study site: 12-Lead ECG to be obtained in triplicate (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.8 Treatment Day 14 (Dose 3)

On Day 14 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)

- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.9 Dose 3 Follow-up Day 19

On Day 19 ( $\pm$  6 hours) the subject may return to the clinic, or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.10 Treatment Day 21 (Dose 4)

On Day 21,  $(\pm 6 \text{ hours})$  subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)

• AE assessment (Section 6.10)

## After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.11 Treatment Day 28 (Dose 5)

On Day 28 ( $\pm$  1 Day), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (collected just prior to the start of the study drug infusion; record collection date and time for each PK sample) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Immune phenotyping
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion

- and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.12 Follow-up Day 29

On Day 29 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.13 Follow-up Day 30

On Day 30 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.14 Follow-up Day 33

On Day 33 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 28), subjects will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.15 Follow-up Day 42

On Day 42 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.16 Follow-up Day 56 (End-of-Study) or Early Termination Visit

On Day 56 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the sitting position) (Section 6.5)
- Serum tetanus antibody and VZV antibody; Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3

- AECA
- RNAseq
- Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.17 Extended Follow-up Visits

Extended follow-up visits will occur only if additional testing for anti-tetanus and/ or anti-VZV titers are required. These visits will occur as needed at approximately 2 months post last dose and 3 months post last dose. See Section 6.7.3.

#### 8 REMOVING SUBJECTS FROM STUDY

Every reasonable effort will be made to keep the subject in the study; however, if a subject is withdrawn from the study, every effort will be made by the Investigator to complete and report the reasons for withdrawal as thoroughly as possible. The reason(s) for termination must be clearly documented on the appropriate page of the eCRF. Once a subject discontinues from the study for any reason, every effort will be made to collect all clinical and laboratory data as scheduled for the Early Termination Visit (See Table 1). A termination eCRF must be completed for all enrolled subjects.

### 8.1 Subject Withdrawal

A subject's participation in the study may be prematurely discontinued for any of the following reasons:

- 1. The subject wishes to withdraw from the study.
- 2. Request by a regulatory agency (e.g., Institutional Review Board).
- 3. Subject experiences a significant or intolerable AE.
- 4. The subject experiences a significant adverse change in vital signs, PE findings, or a clinical laboratory parameter.
- 5. The subject has a need for a concomitant medication that is not permitted by the study protocol.
- 6. The subject experiences generalized impairment or mental incompetence that would result in the subject being unable to understand his or her participation in the study.
- 7. If, in the Investigator's medical judgment, further participation would be injurious to the health and well-being of the subject, or is not in the best interest of the subject.
- 8. Administrative reasons, such as subject non-compliance or a major protocol violation.

Subjects who are withdrawn from this study due to an AE determined to be related to study drug are to be followed until there is either:

- Resolution or stabilization of the AE determined to be related
- The subject is lost to follow-up
- The event is otherwise explained

If there is a persistent AE contributing to discontinuation that is determined to be related to SYNT001, subjects must be followed with appropriate medical management until resolution or stabilization.

A reasonable effort should be made to contact any subject lost to follow-up during the study to complete assessments and retrieve any outstanding data. If the subjects are unreachable by telephone after three (3) attempts, the minimum of a registered letter should be sent requesting that contact be made with the Investigator to report survival information.

#### 8.2 Study Discontinuation

Syntimmune Inc. has the right to terminate or to stop the study at any time. Reasons for study discontinuation may include, but are not limited to the following:

- The incidence or severity of AEs in this or other related studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Drug supply issues
- Excessive subject self-withdrawal
- Significant protocol violations (e.g., violation of eligibility criteria, dosing errors, missing data for study endpoint analysis)

#### 8.3 Replacements

Enrolled subjects withdrawn for a reason other than an AE will be replaced if they have not been dosed or have only received one dose of study drug at the time of discontinuation, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through 28 days after their last dose.

#### 8.4 Stopping Rule

#### 8.4.1 Dose-Escalation Stopping Rule

Dose-limiting toxicity (DLT) will be defined generally as clinically significant, severe (Grade 3) AEs occurring in  $\geq$ 2 subjects that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and no further dose-escalation will occur. If the dose-escalation

stopping rule is met in Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics will be reviewed and a cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met after Cohort 1, dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met in Cohort 2, all safety data and all available pharmacodynamics will be reviewed and a cohort may be added at a dose a minimum of 30% lower than the Cohort 2 dose. If the stopping rule is not met after Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data.

#### 8.4.2 Study Stopping Rule

If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects.

### 8.4.3 Individual Stopping Rule

Dosing for any individual subject will be discontinued (i.e., no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator and Medical Monitor suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject may be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus.

#### 9 STUDY DRUG

For detailed information regarding SYNT001 preparation and administration, refer to the Pharmacy Manual.

#### 9.1 SYNT001

SYNT001 is provided in vials containing 5 mL SYNT001 (extractable volume) at a nominal concentration of 50 mg/mL. The product is supplied as a liquid at pH 6.5  $\pm$  0.5. SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for infusion. SYNT001 will be infused via IV in 250 mL over 1 hour using a 0.2-micron, inline filter.

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these two cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

The specification for host cell DNA in SYNT001 is < 2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing is limited to 5000 mg of SYNT001. Therefore, at the highest dose possible in this study (45 mg/kg), maximum subject weight will be limited to 111 kg.

#### 9.2 **Cohort Dosing**

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. Cohort 2, and Cohort 3 if added, will be dosed per the same schedule

#### 9.3 **Timing of Dosing**

On Days 0, 7, 14, 21, and 28, subjects will receive a 60-minute IV infusion of SYNT001 in the morning. The date and time the dose is administered will be recorded.

#### 9.4 **Identity of Investigational Products**

All supplies of SYNT001 will be supplied by Syntimmune and must be stored refrigerated (2°C to 8°C/36°F to 46°F) in the carton and protected from light, in a securely locked area, accessible to authorized persons only, until needed for dose preparation. Qualified site personnel will

inventory the investigational product received and will maintain records of disposition of the drug, including dates, quantity and use.

#### 9.5 Investigational Product Retention at Study Site

The Investigator (or designee) is responsible for maintaining accurate accountability records of the investigational product throughout the clinical study. All study drug received at the site must be inventoried and accounted for in an accountability log provided by the Sponsor. All dispensing and accountability records will be available for Sponsor review. Study drug accountability will be verified during on-site monitoring visits.

Upon the completion or termination of the study, and upon written authorization from the Sponsor, or its representative, all unused and/or partially used study drug should be returned or destroyed at the investigational site, as specified by Sponsor. It is the Investigator's responsibility to ensure that the Sponsor, or its representative, has provided written authorization that procedures for proper disposal of the study drug have been established, and that appropriate records of the disposal are documented and maintained. No unused study drug may be disposed until fully accounted for by the Sponsor monitor (or designee)

#### 9.6 Warnings and Precautions

**Note:** Subjects must not receive any vaccinations from within 2 weeks of screening until 2 months after the last dose of study drug.

#### 9.6.1 Infusion Reaction

SYNT001 will be given as an IV infusion over 1 hour. As with all mAbs administered by IV infusion, infusion reactions are possible. In nonclinical testing of SYNT001 in NHPs, clinical observations were limited to infusion reactions due to the immunogenicity of SYNT001 in NHPs. These reactions included transient emesis/vomitus which typically occurred within 1 hour of dosing at all dose groups, but only after the third weekly infusion following the development of ADAs. Transient histamine-type responses were noted 30 minutes post-dose in some animals in all dose groups, but only following the third weekly infusion as above. These reactions were consistent with a histamine reaction (decreased activity, periocular swelling, erythema, facial flushing, eyelids partially/completely closed, and/or generalized weakness). With the exception of vomitus/emesis and red skin discoloration associated with injection or blood draw sites, these observations spontaneously resolved within 1-hour post-dose. Subsequent pretreatment with intramuscular diphenhydramine prevented further histamine-type reactions. All doses of SYNT001 were administered by bolus infusion over approximately 5 minutes in the NHP

studies. However, all of the observed infusion reactions (including vomitus/emesis and histamine-type reactions) associated with ADAs are not at all predictive of what may occur in humans [Bugelski 2004, Ponce 2009] and furthermore, are not considered relevant to predicting responses in humans [ICH S6(R1) 2011].

Typically, infusion reactions to monoclonal antibodies observed in human studies develop within 30 minutes to 2 hours after the initiation of drug infusion, although symptoms may be delayed for up to 24 hours. Most are mild in severity, although severe and even fatal reactions can occur.

#### Guidelines for Grading and Management of Allergic or Infusion-Related Reactions

Allergic and/or infusion-related reactions include hypersensitivity reactions and cytokine release syndromes. These reactions are experienced by patients during or within hours of the infusion of monoclonal antibody therapy. Symptoms can include flushing, alterations in heart rate and blood pressure, dyspnea, bronchospasm, back pain, fever, urticaria, edema, nausea, and all types of rashes. Anaphylaxis is recognized as a severe, life-threatening, generalized, or systemic reaction. This is a medical emergency characterized by rapidly developing life-threatening airway and/or breathing and/or circulation problems usually associated with skin or mucosal changes.

Management of Grade 1 infusion reactions include decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen.

Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. See Figure 1 and Figure 2 for details on the management of Grades 1-2 and Grade 3 or higher infusion reactions. The severity of and management of allergic or infusion-related reactions will be graded and managed using NCI CTCAE Version 4.03 (see Table 6).

Figure 1: Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions



If symptoms and signs resolve completely either spontaneously or after administration of diphenhydramine with or without hydrocortisone, consider rechallenge:

Wait at least 20 minutes following medication administration before commencing rechallenge at an infusion rate of 50% or less of the initial infusion rate or

Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction

Figure 2: Management of Severe (Grade 3 or higher) Infusion Reactions

Subject presents with any of the below:

- Urticaria
- Airway threatened by angioedema
- Angioedema: Lip, mouth, facial swelling
- Respiratory compromise wheezing, dyspnea, stridor or hypoxia
   (O2 saturation < 90%)</li>
- BP < 90 mmHg SBP or >30% decrease from patient baseline



Start basic life support:

- High oxygen flow
- On bed, head down, legs up
- Large bore IV cannula, 1 L normal saline STAT
- Initiate vital signs at least every 15 minutes



Consider (under medial direction):

Epinephrine 1:1000

• 0.3 mg (0.3 mL) IM into lateral thigh



Airway Threatened: Nebulized epinephrine 1:1000, 3–5 mL (3–5 mg)

**Bronchospasm:** Nebulized salbutamol 5 mg

(Wheeze or Hypoxia) Consider: Intubation / nebulized epinephrine

**Hypotension:** Place on cardiac monitor

(Systolic BP <100 mmHg) Further epinephrine 1:1000, 0.3 mg IM and

IV normal saline bolus 20 mL/kg STAT as needed

Have vasopressin on hand



Transfer to Emergency Room/ICU Observe until all symptoms resolved.

Table 5: Grading and Management of Allergic or Infusion-Related Reactions

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Infusion-<br>Related<br>Reaction | Mild transient<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Allergic<br>Reaction | Transient<br>flushing or<br>rash, drug<br>fever<br>< 38.0°C.<br>Intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Anaphylaxis | - | - | Symptomatic<br>bronchospasm, with or<br>without urticarial;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Cytokine<br>release<br>syndrome | Mild<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>pressor or<br>ventilator<br>support<br>indicated | Death |

Abstracted from NCI CTCAE Version 4.03.

#### 9.6.2 Potential Immune Effects

An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels after a single dose and further decreases after multiple doses up to a 70% to 80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within normal limits occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.

Given the normal adult range of IgG of 700 to 1600 mg/dL (in some references), with a mean of 1150 mg/dL, a 50% decrease in the mean would be to 575 mg/dL and a 50% decrease from the low end of the normal range of 700 mg/dL would be to 350 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 140 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency [Ameratunga 2013], the levels will be transient. Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to reverse the low IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

An antibody blocking FcRn is expected to also down modulate innate and adaptive immunity and the catabolism of IgG-containing immune complexes (IC). Specifically, it is expected that anti-FcRn will promote the clearance of IgG-containing ICs and the effects of these IC on stimulating innate immune cell production of inflammatory cytokines (e.g., IL-12, interferon-γ, and tumor necrosis factor [TNF]) and inhibit the processing and presentation of antigens contained within IC and thus the antigen-specific activation of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells. Therefore, subjects with pre-existing conditions that are dependent upon IgG antibodies, such as chronic infections (e.g., HIV, HBV or HCV), will be excluded from this study, as will subjects with active infection in general.

SYNT001 administration could decrease the level of protective antibodies from prior vaccinations. Protective antibody levels for tetanus and varicella-zoster virus (chickenpox) are to be tested in accordance with Section 6.7.3.

#### 10 CONCOMITANT MEDICATION AND TREATMENT

All treatments a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications may result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted

Use of the following treatments will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine.
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

In cases in which concomitant medications are used, details to be recorded include the following: medication name, start date and time, stop date and time, dose, route, frequency, and reason for use. The concomitant medication names are to be coded using the World Health Organization

(WHO) Drug Dictionary (WHO-DD March 2013, Type B2 or later) and classified by anatomical therapeutic chemical (ATC) categories.

#### 11 SAFETY

#### 11.1 Safety Parameters

Clinical and laboratory AEs will be graded using the NCI CTCAE; Version 4.03 (See Appendix A).

Subjects will be monitored throughout the treatment and follow-up period for occurrence of AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status, vital sign measurements, and laboratory data (including PD). Safety parameters to be measured/assessed include PEs, vital sign measurements, hematology, serum chemistries, urinalysis, and ECG.

#### 11.2 Adverse Event Definition

An AE is defined as any untoward medical occurrence in a clinical trial subject associated with the use of a drug, whether considered drug related. An AE can be an unfavorable and unintended sign (e.g., an abnormal laboratory value finding), a symptom, or a disease temporally associated with the use of a drug, without judgment as to causality. An AE can arise from use of the drug (e.g., use in combination with another drug) and from any route of administration, formulation or dose, including an overdose. An AE also includes, but is not limited to, any clinically significant worsening of a pre-existing condition. Examples include:

- Any sign, symptom, physical finding, or laboratory result that has worsened in nature, severity or frequency compared to baseline;
- Reactions from an investigational drug, including those occurring because of an overdose, abuse of the study drug, withdrawal phenomena, sensitivity or toxicity;
- Concurrent illness that was not present or worsens in nature, severity, or frequency compared to baseline;
- Injury or accident; and/or
- Exacerbation of a pre-existing condition.

For data collection, all untoward events that occur after informed consent through 28 days after study drug dosing are to be recorded on eCRFs by the investigational site.

While pregnancy alone is not considered as an AE or SAE, any pregnancy complication(s) should be recorded as an AE(s) or SAE(s) (if applicable). Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions (see below). Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. If a female subject becomes pregnant during the conduct of the study, the Investigator must notify the Sponsor according to the procedures provided in Section 11.3.8).

#### 11.3 Evaluating Adverse Events

The Investigator will determine the seriousness, intensity, and causality of an AE associated with the use of the study drug (i.e., events where there is a reasonable possibility that the event may have been caused by the study drug) based on the definitions that follow.

#### 11.3.1 Serious Adverse Events

(Notify Medpace Safety within 24 hours; document on eCRF)

The SAE definition and reporting requirements are in accordance with Title 21 Part Code of Federal Regulations (CFR) 312.32 and the Guidance for Industry and Investigators Safety Reporting Requirements for Investigational New Drug (INDs) and Bioavailability /Bioequivalence Studies.

SAE: An AE is considered "serious" if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:

• <u>Death:</u> This includes any death that occurs while the subject is "on study" as well as any death that occurs within 28 days after study drug administration.

**Note:** Death is an outcome of an AE, and not an AE. The event(s) that caused death (e.g., illness, accident) is the SAE. Death due to any other cause(s) must also be reported as an outcome of the reportable SAE.

• <u>Life-threatening adverse drug event:</u> An AE or suspected adverse reaction is considered "life threatening" if, in the view of either the Investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

#### • Inpatient hospitalization or prolongation of existing hospitalization:

In the absence of an AE, the Investigator should not report hospitalization or prolongation of hospitalization. This is the case in the following situations:

- Hospitalization or prolongation of hospitalization is needed for a procedure required by the protocol
- Hospitalization or prolongation of hospitalization is part of routine procedure followed by study center

- Hospitalization for survey visits or annual physicals
- Hospitalization for observation with release within 24 hours

In addition, a hospitalization planned before the start of the study for a pre-existing condition, which has not worsened, does not count as an SAE.

# • Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

- Congenital anomaly/birth defect
- <u>Important medical event:</u> An event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 11.3.2 Overdose

An overdose is defined as a significant variation from the recommended/scheduled dosage for a product. The dosing for this study will be conducted in a controlled clinical setting and an overdose is not anticipated. However, in the event of an accident, for this study, an overdose of SYNT001 is considered a dose that is two-fold higher than the intended dose for the subject.

#### 11.3.3 Non-Serious Adverse Events

(Document on eCRF)

All other AEs, not fulfilling the previous definitions, are classified as non-serious.

#### 11.3.4 Protocol-Related Adverse Events

AEs that are not test drug related may nevertheless be considered by the Investigator or the Medical Monitor to be related to the conduct of the clinical study. That is, the event may be related to the fact that a subject is participating in the study. For example, a protocol-related AE may be an event that occurs during a screening period or that is related to a procedure required by the protocol.

#### 11.3.5 Assessment of Causality

A medically qualified Investigator must assess the relationship of any AE (including SAEs) to the use of the investigational product, as related or not related, based on clinical judgment and using all available information, and may include consideration of the following factors:

- Possible alternative causes of the AE, including the disease under treatment, pre-existing conditions, concomitant use of other drugs, and presence of environmental or genetic factors
- The temporal association between drug exposure and onset of the AE.
- Whether the manifestations of the AE are consistent with known actions or toxicity of the investigational product.
- The AE resolved or improved with decreasing the dose or stopping use of the investigational product (dechallenge). Judgment should be used if multiple products are discontinued at the same time.

The causal relationship between the study medication and the AE will be assessed using one of the following categories:

**Not Related:** Factors consistent with an assessment of Not Related include:

- Temporal relationship is lacking (e.g., the event did not occur within a reasonable time frame following administration of the study medication); or
- Other causative factors more likely explain the event (e.g., a pre-existing condition, other concomitant treatments).

**Related:** Factors consistent with an assessment of Related include:

• There is a positive temporal relationship (e.g., the event occurred within a reasonable time frame following administration of study medication); or

The AE is more likely explained by the investigational product than by another cause (i.e., the AE shows a pattern consistent with previous knowledge of the investigational product or the class of the investigational product)

#### 11.3.6 Recording Adverse Events

All AEs (including SAEs) are to be accurately recorded on the <u>Adverse Event</u> page of the subject's eCRF. The severity of each AE will be graded using the NCI CTCAE, Version 4.03. The date of onset as well as the end date of the event also should be recorded or the event should be entered as "ongoing". In addition, the method used to treat the AE and the outcome of the AE also will be noted. The Investigator will assess the relationship of the event to study drug.

#### 11.3.7 Planned Hospitalization

A hospitalization planned by the subject prior to the first dose of study medication is considered a therapeutic intervention and not the result of a new SAE and should be recorded as medical

history. If the planned hospitalization or procedure is executed as planned, the record in the subject's medical history is considered complete. However, if the event/condition worsens during the trial, it must be reported as an AE.

#### 11.3.8 Reporting Pregnancies

If a female subject or the female partner of a male subject becomes pregnant during the course of the study, the Investigator must report the pregnancy to the Medpace Safety using the **Pregnancy Reporting Form** within **24 hours** of becoming aware of the event. The Investigator must obtain consent to collect pregnancy information (including the status of the newborn, if applicable).

If some of the information required for completion of the Pregnancy Reporting Form is unavailable at the time of the initial report, follow-up reports will be completed and submitted within 24 hours of becoming aware of the new information. Any pregnancy will be followed through delivery for the observation of any SAEs. Any SAE that occurs during pregnancy must be recorded on the SAE report form in the EDC system (e.g., maternal serious complications, therapeutic or spontaneous abortion, ectopic pregnancy, stillbirth, neonatal death, congenital abnormality, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs (See Section 11.3.9).

#### 11.3.9 Serious Adverse Event Reporting

#### 11.3.9.1 Governing Regulatory Requirements

Compliance with this request for prompt reporting is essential in that the sponsor is responsible for informing the US Food and Drug Administration (FDA) and other regulatory authorities as well as all other participating Investigators of the event.

Under FDA ruling (US Code of Federal Regulations, Title 21 CFR Part 312.32) and the ICH Guidelines for Clinical Safety Data Management Definitions and Standards for Expedited Reporting, the sponsor is required to submit written documentation, in the form of a safety report, detailing:

- Any event associated with the use of the drug, that is both serious and unexpected, or
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects, including reports of mutagenicity, teratogenicity, or carcinogenicity.
Written submission must be made by the sponsor to the FDA and the IRBs as soon as possible and in no event later than 15 calendar days after the sponsor's initial notification of the event. The sponsor shall also inform all Investigators.

#### 11.3.9.2 Time Frame for Reporting

Any death, SAE, pregnancy, or unexpected (and severe) AE experienced by the subject after informed consent or within 28 days of receiving study drug, regardless of relationship to study drug, or any death that occurs more than 28 days after receiving study drug, and is believed to be study drug related, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee).

Contact information for **SAE** reporting:



Additionally, the Investigator will be able to contact the **Medical Monitor**:



#### 11.3.9.3 Information to be Provided by the Investigator

SAEs must be recorded on the SAE form in the EDC system. This requirement includes all SAEs that occur after informed consent and through 28 days after study drug dosing, and in addition, any SAE that are assessed as related to study treatment by the Investigator, even if the SAE occurs more than 28 days after study drug dosing.

The minimum information required for SAE reporting includes identity of Investigator, site number, subject number, an event description, SAE term(s), onset date, the reason why the event is serious (i.e., the seriousness criteria) and the Investigator's assessment of the relationship of the event to study treatment. Additional SAE information including medications or other therapeutic measures used to treat the event, action taken with the study treatment due to the event, and the outcome/resolution of the event will be recorded. Paper forms for reporting SAEs will be provided to the study sites as back-up in case the EDC system is not accessible.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. Furthermore, the Investigator may be required to provide supplementary information as requested by Syntimmune or designee.

When reporting an SAE, the following additional points should be noted:

When the diagnosis of an SAE is known or suspected, the Investigator should report the diagnosis or syndrome as the primary SAE term, rather than as signs or symptoms. Signs and symptoms may then be described in the event description. For example, dyspnea should not be used as an SAE term if the diagnosis, which caused the dyspnea, is known to be malignant pleural effusion.

- Death should not be reported as an SAE, but as an outcome of a specific SAE, unless the event preceding the death is unknown. In the exceptional case where the events leading to death are unknown, then death may be used as an event term. If an autopsy was performed, the autopsy report should be provided.
- While most hospitalizations necessitate reporting of an SAE, some hospitalizations do not require SAE reporting, as follows:
  - Elective or previously scheduled surgery, e.g., a previously scheduled ventral hernia repair
  - Procedures for pre-existing conditions that have not worsened after initiation of treatment
  - Pre-specified study hospitalizations for observation
  - Events that result in hospital stays of less than 24 hours and that do not require admission, e.g., an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics
- SAEs must, however, be reported for any surgical or procedural complication resulting in prolongation of the hospitalization.

#### 11.3.10 **Regulatory Reporting**

Syntimmune (or designee) will process and evaluate all SAEs as soon as the reports are received. For each SAE received, Syntimmune will decide as to whether the criteria for expedited reporting have been met.

Syntimmune (or designee) will submit SAEs that meet the criteria for expedited reporting to the regulatory authorities in accordance with local regulations governing safety reporting. Reporting of SAEs by the Investigator to his or her IRB will be done in accordance with the standard operating procedures and policies of the IRB. Adequate documentation must be maintained showing that the IRB was properly notified.

#### 11.3.11 Follow-up Information on a Serious Adverse Event (SAE)

Appropriate diagnostic tests should be performed and therapeutic measures, if indicated, should be instituted. Appropriate consultation and follow-up evaluations should be carried out until the event has returned to baseline or is otherwise explained by the Investigator.

If all required information on the SAE form is not available at the time of the initial report, follow-up information will be completed in the EDC system.

#### 11.4 Other Safety Considerations

#### 11.4.1 Laboratory Data

All laboratory data obtained during the study should be reviewed. Any abnormal value that leads to a change in subject management (e.g., requirement for additional medication or monitoring) or is of clinical significance by the Investigator should be reported as an AE and/or SAE as appropriate, unless this value is consistent with values obtained before entry into the study.

#### 11.4.2 Medication Errors

Any medication error that results in an AE, even if it does not meet the definition of serious, requires reporting within 24 hours to the safety Medical Monitor.

#### 11.4.3 Follow-Up of Adverse Events

Any SAE or AE assessed as related that led to treatment discontinuation (including clinically significant abnormal laboratory values that meet these criteria) and ongoing 28 days after study drug dosing must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. This follow-up guidance also applies to related SAE that occur more than 28 days after study drug dosing. The status of all other continuing AEs will be documented as of 28 days after study drug dosing. The Investigator will follow all subjects who experience AEs until there is a return to the subject's baseline condition, or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary.

Where a diagnosis is possible, it is preferable to report this diagnosis rather than a series of terms (signs/symptoms) relating to the diagnosis.

#### 11.5 Safety Monitoring for Dose Escalation

Following dosing in each cohort, all safety/tolerability data (e.g., PEs, vital signs [including pulse oximetry], clinical safety laboratory tests, ECGs and AE/SAE assessments) as well as any available and relevant PD data collected through Day 42 will be reviewed by the DEC. A decision to escalate to the next cohort will be made. The recommendation may be to continue to the next scheduled dose level, discontinue the study or to modify dosing to a dose less than the current dose or higher than the current dose but lower than the next planned dose.

#### 12 STATISTICAL CONSIDERATIONS

All descriptive and inferential statistical analyses will be performed using the most recently released and available Statistical Analysis System (SAS) software, unless otherwise noted. Missing data will not be imputed unless otherwise stated. All clinical data captured will be provided in data listings. A Statistical Analysis Plan (SAP) and a Pharmacokinetic Analysis Plan (PAP) will be finalized prior to database lock.

#### 12.1 General Design

All data for enrolled subjects will be presented in data listings by subject number.

Continuous data will be described using descriptive statistics: number of observations (n), mean, standard deviation (SD), median, minimum, and maximum. Frequencies and percentages will be used for summarizing discrete (categorical) data. When categorical data are presented, the percent will be suppressed when the count is zero to draw attention to the non-zero counts. The denominator for all percentages, unless otherwise specified, will be the number of subjects in the specified analysis population.

#### 12.2 Sample Size Justification

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

#### 12.3 Statistical Considerations

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). The SAP may modify the plans outlined in the protocol; any deviations from the previously described statistical plan will be described and justified in an SAP amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate and will be described in the SAP. Methods of handling of missing data for different endpoints will be further specified in the SAP. In general, where individual data points are missing because of insufficient samples, dropouts, or other reasons, the data will be analyzed based on reduced denominators unless specified otherwise in the SAP.

Results will be summarized by cohorts.

#### 12.3.1 Study Populations

Three populations will be employed in the analysis of study data:

- The **intent-to-treat (ITT)** population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population.
- The **PK** population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters.
- The **PD** population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the ITT, PK, and PD populations, where appropriate.

#### 12.3.2 Subject Accountability, Demographics, and Baseline Characteristics

Subject disposition, demographic information and baseline characteristics will be presented. Any discrepancy between treatment to be given and treatment received will be accounted for in these displays.

#### 12.3.3 Concomitant Medications

Concomitant medications will be coded using WHO Drug Dictionary (WHO-DD March 2013, Type B2 or later) and the data will be summarized and presented in tables and listings.

#### 12.4 Planned PK Analysis

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and  $AUC_{0-24}$  and  $AUC_{0-\infty}$ . PK parameters will be determined using noncompartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, SD, coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

For calculation of mean concentrations and generation of mean concentration-time profiles, all below the limit of quantification (BLQ) values will be set to zero except when an individual BLQ falls between 2 quantifiable values, in which case it will be omitted.

If there are values above the BLQ, but too sparse to allow full analysis, descriptive statistics will be performed on available values.

### 12.5 Safety Data

Safety observations and measurements include AEs, safety laboratory tests, vital sign measurements, PEs, and ECGs.

Treatment-emergent AEs will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

AEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject, cohort, and overall per SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by cohort. Incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the local laboratory.

Vital sign measurements and change from baseline will be summarized at each scheduled time point by cohort using descriptive statistics.

Arithmetic mean of parameters from triplicate ECG will be calculated first for each participant at each planned time point. Then summary statistics of ECG test parameters (mean of triplicate) and change from baseline to each post-dose time point will be calculated. Shift tables for ECG test result category change (normal, abnormal, clinically abnormal) from pre-dose to each post-dose time point showing number and percentage of subjects with movement between categories will be presented by treatment group. Frequency and percentage of subjects experiencing potential QTc prolongation (QTcF > 450) will be summarized at each time point by cohort.

#### 12.6 Pharmacodynamic/Activity Data

PD results will be summarized by cohort.

#### 12.7 Immunogenicity Data

Immunogenicity results will be summarized by cohort.

# 12.8 Interim Analysis

No interim analysis is planned. Safety results will be examined for making dose-escalation decisions; no statistical analyses are planned for aiding these dose-escalation decisions.

#### 13 DATA QUALITY ASSURANCE

All data will be entered in a validated electronic data capture system using single data entry. Standard procedures (including following data review guidelines, manual clinical review based on subject profiles, computerized validation to produce queries, and maintenance of an audit file which includes all database modifications) will be followed to ensure accurate data. Clinical personnel will review all data listings for outliers, data inconsistencies, and spelling errors.

During the study, a study site monitor will make site visits to review protocol compliance, compare electronic case report forms (eCRFs) against individual subject medical records, assess drug accountability, and ensure that the study is being conducted using pertinent regulatory requirements. eCRF entries will be verified with source documentation. The review of medical records will be performed in a manner to ensure that subject confidentiality is maintained. Checking the eCRFs for completeness, clarity and cross checking with source documents is required to monitor the progress of the study. Direct access to source data is also required for inspections and audits, and will be carried out giving due consideration to data protection and medical confidentiality. Each Investigator will have assured Syntimmune of full access to complete source data for study participants and associated necessary support at all times.

In addition to routine monitoring procedures, audits of clinical research activities in accordance with standard operating procedures (SOPs) may be performed to evaluate compliance with the principles of GCP. A regulatory authority may also wish to conduct an inspection (during the study or even after its completion). If a regulatory authority requests an inspection, the Investigator must immediately inform Syntimmune that this request has been made. Study conduct may be assessed during the study by a Clinical Quality Assurance representative(s) to ensure that the study is conducted in compliance with the protocol. This designee, as well as the site monitor, will be permitted to inspect the study documents (study protocol, eCRFs, investigational product accountability, original study-relevant medical records). All subject data will be treated confidentially. During the clinical study, access will be available to Syntimmune or their designee (e.g., contract research organization [CRO]) to view the eCRFs after completion of the individual sections of the study. Furthermore, the study protocol, each step of the data-recording procedure and the handling of the data as well as the study report may be subject to independent review by a Quality Assurance representative. Clinical site and study audits will be conducted as necessary to assure the validity of the study data.

#### 14 STUDY ADMINISTRATION

#### 14.1 Study Administrative Structure

The study administration structure is provided in Table 6.

**Table 6:** Study Administrative Structure



#### 14.2 Ethical Conduct of the Study

The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH E6 Tripartite Guideline (January 1997), and in general, be conducted in a manner consistent with the principles described in the Declaration of Helsinki. The Investigator will ensure that the conduct of the study complies with the basic principles of GCP as outlined in the current version of 21 CFR, subpart D, Part 312, "Responsibilities of Sponsors and Investigators", Part 50, "Protection of Human Subjects", and Part 56, "Institutional Review Boards".

#### 14.3 Informed Consent (ICF)

A properly executed, written informed consent document, in compliance with 21 CFR, Part 50 and the ICH guidelines, will be obtained from each subject before the subject is entered into the study and before any study screening procedure is performed that involves risk. Attention will

be directed to the basic elements required for incorporation into the informed consent under US Federal Regulations for Protection of Human Subjects (21 CFR 50.25[a]) and (21 CFR 50.25[b]), as necessary.

Sample ICFs will be supplied to each site. Syntimmune or its designee must review any proposed deviations from the sample ICF. The final IRB-approved document must be provided to Syntimmune for regulatory purposes.

It is the responsibility of the Investigator, or a person designated by the Investigator, to obtain written informed consent from each subject (or the subject's legally authorized representative) participating in this study after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study. In the case where the subject is unable to read, an impartial witness should be present during the entire informed consent discussion. After the subject has orally consented to participation in the trial, the witness' signature on the form will attest that the information in the consent form was accurately explained and understood. A copy of the ICF must be provided to the subject or to the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

The eCRF for this study contains a section for documenting informed subject consent, and this must be completed appropriately. Signed ICFs must remain in each subject's study file and must be available for verification by site monitors at any time. If new safety information results in significant changes in the risk/benefit assessment, the consent form should be reviewed and updated as necessary. All subjects (including those already being treated) should be informed of the new information, should be given a copy of the revised form, and should give their consent to continue in the study.

#### 14.4 Institutional Review Board

This study is being conducted under US IND 128152. This protocol (and any modifications) and appropriate consent procedures must be reviewed and approved by an IRB. This board must operate in accordance with the current federal or local regulations. The Investigator will send a letter or certificate of IRB approval to Syntimmune (or designee) before subject enrollment and whenever subsequent modifications to the protocol are made.

#### **14.5 Dose Escalation Committee**

The DEC will be responsible for confirming the safety of the investigative product prior to dose escalation, as well as the dose level for each successive cohort. In addition, over the course

of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects. The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions.

#### 14.6 Future Use of Subject Samples

Not all the tissue and blood components obtained during this study may be required for the tests that are part of the clinical trial. Available samples may be used for additional research. This research will help to understand disease subtypes, drug response and AE, and possibly identify new drug targets or biomarkers that predict subject response to treatment. The use of the samples for internal research will be done using the guidelines defined by the FDA guidance for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individual Identifiable (issued 25 April 2006) and the European Medicines Agency (EMA) Reflection Paper on Pharmacogenetic Samples, Testing and Data Handling (Doc. Ref.

EMEA/CHMP/PGxWP/201914/2006; 15 November 2007). If a subject requests destruction of their tissue and blood samples and the samples have not yet been de-identified, Syntimmune will destroy the samples as described in this FDA guidance. Syntimmune will notify the Investigator in writing that the samples have been destroyed.

#### 15 CONDITIONS FOR MODIFYING THE PROTOCOL

Protocol modifications to ongoing studies must be made only after consultation between a Syntimmune representative and the Investigator. Protocol modifications will be prepared, reviewed, and approved by Syntimmune representatives.

All protocol modifications must be submitted to the IRB for information and approval in accordance with local requirements, and to regulatory agencies if required. Approval must be obtained before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to study subjects, or when the change involves only logistical or administrative aspects of the trial (e.g., change in site monitor, change of telephone number).

#### 16 CONDITIONS FOR TERMINATING THE STUDY

Syntimmune has the right to terminate the study at any time. In terminating the study, Syntimmune and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests.

#### 17 STUDY DOCUMENTATION, CRFS, AND RECORD KEEPING

#### 17.1 Investigator's Files and Retention of Documents

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into 2 separate categories as follows: (1) Investigator's study file and (2) subject clinical source documents.

The Investigator's study file will contain the protocol and protocol amendments, eCRFs, query forms, IRB and governmental approval with correspondence, sample informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

Subject clinical source documents (usually predefined by the project to record key efficacy and safety parameters independent of the eCRFs) may include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, electroencephalogram, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject screening and enrollment logs. The Investigator must keep these 2 categories of documents on file for at least 2 years following the marketing application approval date for the study treatment and for the indication being investigated or for 2 years after the development program is discontinued and the FDA notified. After that period, the documents may be destroyed subject to local regulations with prior written permission from Syntimmune. If the Investigator wants to assign the study records to another party or move them to another location, Syntimmune must be notified in advance.

If the Investigator cannot guarantee the archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and Syntimmune to store these in a sealed container outside of the study site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storing outside of the study site.

#### 17.2 Source Documents and Background Data

Investigators must maintain adequate and accurate source documents on which the eCRFs for each subject are based. They are separate and distinct from the eCRFs.

These records include detailed notes on the following:

Syntimmune, Inc.

- Medical history
- Date and time of informed consent with Health Insurance Portability and Accountability
  Act (HIPAA) authorization either contained in the ICF or presented to the subject
  candidate as a standalone document
- Description of the complete consenting process
- The basic identifying information that linked the subject's medical record with the eCRFs
- The results of all diagnostic tests performed, diagnoses made, therapy provided, and any other data on the condition of the subject
- The medical condition of the subject during their involvement in the study
- All AEs
- The subject's exposure to the study medication
- The subject's exposure to any concomitant therapy
- All relevant observations and data on the condition of the subject throughout the trial
- Justification for all entries in the subject's eCRF

A subject log of all potentially eligible subjects considered, but not consented, for obvious deviations from the entry criteria, will be kept at each site. The log will contain subjects' initials, diagnosis, eligibility, or, if not eligible, reason for not consenting. All consented subjects will be logged, regardless of whether they ultimately enroll.

Upon request, the Investigator will supply Syntimmune with any required background data from the study documentation or clinic records. This is particularly important when eCRFs are illegible or when errors in data transcription are suspected. In case of special problems or governmental queries or requests for audit inspections, it is also necessary to have access to the complete study records, provided that subject confidentiality is protected.

#### 17.3 Audits and Inspections

The Investigator should understand that source documents for this study should be made available to appropriately qualified personnel from Syntimmune (or designee), or to health authority inspectors after appropriate notification. The verification of the eCRF data must be by direct inspection of source documents.

#### 17.4 Electronic Case Report Forms

Clinical trial data for this study will be captured on eCRF designed for computer processing and analysis. This computerized system will be validated and compliant with 21 CFR Part 11. Corrections to data will be made using 21 CFR Part 11, Electronic Records; Electronic Signatures. If corrections are made after review and sign-off by the Investigator, he/she must be aware of the changes and provide written acknowledgement. There will also be an electronic audit trail. Corrections on paper CRFs must be initialed and dated by the person making the change. The Investigator agrees to provide all information requested on the eCRF in an accurate manner using instructions provided. The Investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported to Syntimmune in the eCRF and in all required reports.

An eCRF is required to be submitted for every subject who receives any amount of study drug. This includes submission of retrievable data on subjects who withdraw before completion of the study. Prior to submission, eCRFs must be reviewed for completeness and accuracy, and signed and dated where either indicated, by the Principal Investigator or authorized delegate from the study staff. If a subject stops treatment or terminates from the study, the dates and reasons must be noted on the eCRF.

#### 18 MONITORING THE STUDY

It is understood that the responsible Syntimmune site monitor (or designee) will contact and visit the Investigator regularly and will be allowed on request to inspect the various records of the trial (eCRFs and other pertinent data) if subject confidentiality is maintained in accordance with local requirements.

It will be the site monitor's responsibility to inspect the eCRFs at regular intervals throughout the study, to verify the adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The site monitor should have access to laboratory test reports and other subject records needed to verify the entries on the eCRF. The Investigator (or designee) must agree to cooperate with the site monitor to ensure that any problems detected during these monitoring visits are resolved.

#### 19 CONFIDENTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECORDS

The Investigator must ensure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On eCRFs or other documents submitted to Syntimmune, subjects should be identified by an identification code and not by their names. The Investigator should keep a subject enrollment log showing codes, names, and addresses. The Investigator should maintain documents not for submission to Syntimmune (e.g., subjects' written consent forms) in strict confidence.

Authorized regulatory officials and Syntimmune personnel (or their representatives) will be allowed full access to inspect and copy the records. All study drugs, subject bodily fluids and tissue, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by Syntimmune.

The Principal Investigator also agrees that all information received from Syntimmune, including but not limited to the IB, this protocol, eCRFs, the INDs, and any other study information remain the sole and exclusive property of Syntimmune during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from the sponsor. The Principal Investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 20 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. The Investigator agrees that any manuscript or abstract they author may be published only after receiving written permission from Syntimmune.

If Syntimmune coordinates a publication or presentation of study results from all study sites, the participation of Investigator or other representatives of study site as a named author shall be determined in accordance with Syntimmune policy and generally accepted standards for authorship.

#### 21 REFERENCES

Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID), which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. *Clin. Exp. Immunol.* 2013;174: 203-211.

Bugelski PJ and Treacy G. (2004) Predictive power of preclinical studies in animals for the immunogenicity of recombinant therapeutic proteins in humans. *Curr Opin Mol Ther*. 2004;6:10–16.

International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) (2011). S6(R1) Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals. Accessed 03 June 2016.

http://www.ich.org/products/guidelines/safety/safety-single/article/preclinical-safety-evaluation-of-biotechnology-derived-pharmaceuticals.html

Nixon AE, Chen J, Sexton DJ, Muruganandam A, Bitonti AJ, Dumont J, Viswanathan M, Martik D, Wassaf D, Mezo A, Wood CR, Biedenkapp JC, TenHoor C. (2015). Fully human monoclonal antibody inhibitors of the neonatal Fc receptor reduce circulating IgG in non-human primates. Front. Immun. 6:176

Ponce R, Abad L, Amaravadi, L, et al. Immunogenicity of biologically-derived therapeutics: assessment and interpretation of nonclinical safety studies. *Regul Toxicol Pharmacol*. 2009;54,164–182.

Roopenian, D.C., Christianson, G.J., Sproule, T.J., Brown, A.C., Akilesh, S., Jung, N., Petkova, S., Avanessian, L., Choi, E.Y., Shaffer, D.J., Eden, P.A., Anderson, C. L. The MHC class I-like IgG receptor controls perinatal IgG transport, IgG homeostasis, and fate of IgG-Fc-coupled drugs. 2003. J. Immun. 170 3528-3533

Appendix A: NCI CTCAE, Version 4.03

# Appendix B: Pemphigus Disease Area Index (PDAI)

# Pemphigus Disease Area Index (PDAI)

| Skin | Activity | | Damage |
|---|---|---|---|
| Anatomical Locatio | Erosion/Blisters or new erythema | | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion |
| | 0 absent 1 1-3 lesions, up to one >2 cm in any diameter, none > 6 cm 2 2-3 lesions, at least two > 2 cm diameter, none > 6 cm 3 >3 lesions, none > 6 cm diameter 5 >3 lesions, and/or at least one >5 cm diameter of cm diameter of cm diameter of cm diameter or entire area | | 0 absent<br>1 present |
| Ears | | | |
| Nose | | | |
| Rest of the face | | | |
| Neck | | | |
| Chest | | | |
| Abdomen | | | |
| Back, buttocks | | | |
| Arms | | | |
| Hands | | | |
| Legs | | | |
| Feet | | | |
| Genitals | | | |
| Total skin | /120 | | /12 |
| Scalp | | | |
| Scalp | Erosion/Blisters or new erythema | | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion |
| | 0 absent 1 in one quadrant 2 two quadrants 3 three quadrants 4 affects whole skull 10 at least one lesion > 6 cm | | 0 absent<br>1 present |
| Total Scalp (0-10) | /10 | | /1 |
| Mucous mer | nbrane | | 1 |
| Anatomical<br>Location | Erosion/Blisters | | |
| | 0 absent<br>1 1 lesion<br>2 2–3 lesions<br>5 >3 lesions or 2 lesions >2 cm<br>10 entire area | Number<br>lesions<br>if ≤ 3 | |
| Eyes | | $\sqcup$ | |
| Nose | | $\sqcup$ | |
| Buccal mucosa | | | |
| Hard palate | | $\vdash$ | |
| Soft palate | | $\vdash$ | |
| Upper gingiva | | $\vdash$ | |
| Lower gingiva | | $\vdash$ | |
| Tongue | | $\vdash$ | |
| Floor of mouth | | $\vdash$ | |
| Labial bucosa | | $\vdash$ | |
| Posterior pharynx | | <del> </del> | |
| | /120 | | |

Copyright ©2007 University of Pennsylvania; All Rights Reserved.

# Syntimmune, Inc.

#### SUMMARY OF CHANGES TO CLINICAL STUDY PROTOCOL

A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

**Medical Monitor:** PPD

43 Thorndike Street, Cambridge, MA 01240

Phone: PPD extension PPD

Mobile: PPD

Original Protocol: 28 January 2017 Amendment 1.1 21 March 2017

#### **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

#### **SUMMARY**

The SYNT001-103 protocol has been amended with administrative changes as follows:

- Removal of Anti-desmoglein (1&3) antibody testing on Day 28 from the Study Assessments table.
- Total blood draw for subjects completing the study at Day 56 updated to approximately
   311 mL in Section 6.7
- Corrected format and reference for the Pemphigus Disease area Index (PDAI) in Appendix B

#### **SPECIFIC CHANGES**

Text deletions are shown using strike through font; additions in *italic font*.

#### **SECTION 1, STUDY SYNOPSIS**

**Table 1, Study Assessments** 

**Anti-Dsg (1&3) antibody titer:** 'X' removed from Day 28 box. Incorrectly included in the Study Assessments Table.

#### **SECTION 6 STUDY PROCEDURES**

#### **Section 6.7, Clinical Laboratory Measurements**

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and anti-drug antibody samples) will be performed using established methods by a central laboratory. Safety laboratory panels are defined as listed in Table 3. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and anti-drug antibody samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42 and 56. The total blood draw for each subject who completes the study at Day 56, will be approximately 308 311 mL. Please refer to the Laboratory Manual for more information

#### **APPENDIX B:**

#### Pemphigus Disease Area Index (PDAI)

Replaced PDAI form with an updated version as provided by University of Pennsylvania

# Syntimmune, Inc.

#### **CLINICAL STUDY PROTOCOL**

# A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

**Medical Monitor:** PPD

43 Thorndike Street, Cambridge, MA 01240

Phone: PPD extension PPD

Mobile: PPD

Original Protocol:18 January 2017Amendment 1.1:21 March 2017Amendment 2.012 April 2017

#### **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

#### **SPONSOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the Investigator, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| PPD | |
|-----|-------------------|
| | 13-4-2017 |
| | Date of Signature |
| | (DD Mm YYYY) |

#### PROCEDURES IN CASE OF EMERGENCY

#### Serious Adverse Events

Any death, serious adverse event (SAE)\* occurring in a subject while receiving study drug or within 7 days of receiving study drug, even though the event may not appear to be study drug related, must be promptly reported (within 24 hours) by telephone or electronic communication to the sponsor (or designee).

#### **Emergency Contact Information**

| For SAE reporting: | | For any other questions or to contact the Medical Monitor: |
|---|---|---|
| Medpace Clinical Safety | | PPD |
| Medpace SAE hotline: | | PPD |
| Telephone: PPD | dial P or PPD | Mobile phone: PPD Office phone: PPD ext. PPD |
| PPD dial P | D | Office phone: PPD ext. PPD |
| Facsimile: PPD | or PPD | |
| PPD | | |

#### **SAE CRITERIA**

- \* A <u>serious adverse event</u> (SAE) is any untoward medical occurrence that at any dose results in any of the following outcomes, regardless of relationship to study drug (see Section 11.3.1, Serious Adverse Events for additional information):
  - Death
  - Life-threatening adverse drug event
  - Inpatient hospitalization or prolongation of existing hospitalization
  - A persistent or significant disability/ incapacity
  - A congenital anomaly/birth defect
  - An important medical event that may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

Syntimmune, Inc.


Amendment 2.0 Final 12 April

#### **INVESTIGATOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the sponsor, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonization Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

Nothing in this document is intended to limit the authority of a physician to provide emergency

| medical care under applicable regulations. | |
|--------------------------------------------|--------------------------------|
| Investigator Signature | Date of Signature (DD Mm YYYY) |
| Name of Investigator (please print) | |

#### 1 SYNOPSIS

| Study title | A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus) |
|---|---|
| Protocol number | SYNT001-103 |
| Number of study centers | Approximately 10 (US) |
| Clinical phase | Phase 1b |
| Study background | SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG immune complexes from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG containing immune complexes further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG immune complexes within and among compartments important in cellular immunity, it is further anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8+ and CD4+ T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG and IC that are involved in many autoimmune conditions and dismantle their ability to cause disease. SYNT001 targets mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP). While current treatments for certain autoimmune disorders including chronic steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are frequently associated with significant adverse effects, a |

Protocol SYNT001-103

| Study rationale | pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, leading to a significant decrease in total IgG, and thereby a corresponding decrease in the level of the pathogenic autoantibodies as well as the ICs to which they are associated, should lead to a decrease in the mucosal and cutaneous manifestations in subjects with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification. This study is being conducted to further evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity |
|---|---|
| | markers. |
| Study objectives | Primary objective To evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus) |
| | Secondary objectives |
| | <ul> <li>To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels</li> <li>To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers: <ul> <li>Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM</li> <li>Albumin</li> </ul> </li> </ul> |
| | • To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers: |
| | <ul> <li>Serum anti-desmoglein (Dsg) (1 and 3) antibody levels</li> <li>Pemphigus Disease Area Index (PDAI)</li> </ul> |
| | To assess immunogenicity (anti-SYNT001 antibodies) |
| | Exploratory objectives |
| | • To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including: |
| | <ul> <li>Serum anti-epithelial cell antibody (AECA) levels by indirect<br/>immunofluorescence</li> </ul> |
| | <ul> <li>Circulating immune complexes (CIC)</li> </ul> |
| | o Complement component 3 (C3) |
| | <ul> <li>Exploratory biomarkers (FCGR2A (single nucleotide polymorphism-<br/>SNP), RNAseq, urine IgG)</li> </ul> |

# Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells SYNT001 levels in skin biopsies (optional)

- To characterize corticosteroid use during the study

#### Study design

Phase 1b, multicenter, open-label, safety, tolerability, and activity study

#### Methodology

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of subjects | Dose |
|--------|-----------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs, and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All safety data and any available and relevant PD data through Day 42 (2 weeks after the last subject's last dose in Cohort 1) will be reviewed by a dose escalation committee before Cohort 2 is initiated. Escalation to Cohort 2 will proceed if there are no concerning safety signals and the review of available and relevant PD data supports advancing to a higher dose. The dose for Cohort 2 will be finalized after review of the safety and PD data, but will not exceed 30 mg/kg. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule as Cohort 1.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84 and 112. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42 and 56 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, adverse event (AE) assessments, concomitant medication assessments, and electrocardiograms (ECG).

#### **Number of subjects**

Approximately 16; two cohorts of 8 subjects each. An additional cohort of up to 8 subjects may be enrolled. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects with pemphigus foliaceus may be enrolled.

# Diagnosis and main entry criteria

#### **Inclusion criteria:**

Subjects must meet the following criteria to be included:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq 18$  years of age at the time of screening;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal;
  - c. History of at least one positive tissue-based test (e.g., biopsy, direct immunofluorescence [DIF])
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose
     12 months prior to screening;

- b. If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
- c. If being treated with corticosteroids, must be  $\leq 1 \text{mg/kg/day}$  and stable (< 10% change in dose) for 2 weeks prior to screening;
- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 35.0 \text{ kg/m}^2$ ;
- 6. Has a negative urine pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through the final study visit.

#### **Exclusion criteria:**

Subjects meeting any of the following criteria are to be excluded:

- 1. Subject unable or unwilling to comply with the protocol;
- Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG use within 60 days of screening;
- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;
- 8. Any exposure to an investigational drug or device within the 30 days prior to screening
- Plasmapheresis or immunoadsorption within 60 days of screening
| | <del>-</del> |
|---|---|
| | 10. Cellular therapy at any time prior to screening |
| | 11. Use of any immunosuppressive drugs apart from corticosteroids, |
| | azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of |
| | screening |
| | 12. Serum total IgG < 600 mg/dL; |
| | 13. Subject has any current medical condition that, in the opinion of the |
| | Investigator, may compromise their safety or compliance, preclude |
| | successful conduct of the study, or interfere with interpretation of the results |
| | (e.g., a significant pre-existing illness or other major comorbidity that the |
| | Investigator considers may confound the interpretation of the study results); |
| | 14. Any vaccination within 2 weeks of screening |
| Study drug, dosage, | SYNT001 |
| and administration | <b>Doses:</b> 10 mg/kg and 30 mg/kg. A third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive. |
| | SYNT001 is provided as a liquid at a nominal concentration of 50 mg/mL. SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for |
| | infusion. |
| | Route of administration: IV in 250 mL over 1 hour |
| Control, dose, and | Not applicable |
| route of | |
| administration | |
| <b>Duration of subject</b> | Up to 126 days (18 weeks): Screening of up to 2 weeks (14 days); Treatment |
| participation and | period of 8 weeks (56 days); Follow-up period of 8 weeks (56 days) |
| duration of study | |

# Prohibited Concomitant treatments

All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted.

Use of the following medications will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations through Day 56. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator.

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

#### Safety assessments

Safety assessments include AEs, serious adverse events (SAEs), PEs, vital sign measurements, clinical safety laboratory evaluations, ECGs, and reasons for treatment discontinuations due to toxicity. Safety assessments will be performed at specified time points and prior to discharge from the clinic. Vital sign measurements, including blood pressure, pulse rate, respiratory rate, and temperature will be monitored throughout the study. Pulse oximetry will be monitored during the study drug infusion and for 2 hours following the end of the infusion.

The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03) will be used for grading clinical and laboratory AEs.

| | The AE reporting period for a subject enrolled in the study begins when the subject provides informed consent and is continued through the last study visit. All AEs that occur in the enrolled subjects during the AE reporting period must be recorded, regardless of the relationship of the AE to study drug. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug should also be recorded. |
|---|---|
| Dose-escalation rules | Dose escalation decisions will be made by a Dose Escalation Committee (DEC) and will be based on safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities, AEs, SAEs, and total IgG levels. Dose-limiting toxicity (DLT) will be defined generally as severe (Grade 3) AEs occurring in $\geq 2$ subjects that are determined to be clinically significant and considered related to study drug. |
| | If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. If the dose-escalation stopping rule is met during Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics data will be reviewed and the cohort may resume (if applicable) or a new cohort may be added, at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met in Cohort 1 (10 mg/kg), dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met for the first time during Cohort 2, all safety data and all available pharmacodynamics data will be reviewed and the cohort may resume (if applicable) or a new cohort may be added at a dose at least 30% lower than the Cohort 2 dose. If the stopping rule is not met in Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data. |
| Study stopping rule | If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, any further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the next appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects. |
| Individual stopping<br>rule | Dosing for any individual subject will be discontinued (i.e., further treatment with the study drug will not be given) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject will be discontinued from further treatment with |

| | study drug, at the discretion of the Investigator with consultation with the |
|---|---|
| | Medical Monitor, if they require a significant increase in dose(s) of anti- |
| | pemphigus medication(s) for the management of pemphigus. |
| Pharmacokinetics | The PK of SYNT001 will be evaluated following the first and last (fifth) doses of SYNT001. |
| | Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. Study drug concentration will be used to calculate the following PK parameters: $t_{1/2}$ , $C_{max}$ , $T_{max}$ , $AUC_{0-24}$ , and $AUC_{0-\infty}$ . |
| Pharmacodynamics/<br>Activity | PD samples will be collected for analysis of IgG (serial assessment of IgG levels to identify C <sub>min</sub> , T <sub>min</sub> ); IgG1-4 subtype levels; IgA levels; IgM levels; albumin levels; anti-Dsg (1 and 3) antibody levels; serum AECA by direct immunofluorescence; CIC; C3; exploratory biomarkers ( <i>FCGR2A</i> SNP, RNAseq, urine IgG, CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T, monocytes, NK cells and B cells). |
| Immunogenicity | Samples will be collected for immunogenicity analyses on Days 0 (pre-dose), 14, 28, 56, 84 and 112. |
| Skin biopsy | Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33, 56 and 84 to analyze SYNT001 levels. |
| Photography | Photographs of active lesions will be taken at Day 0. Follow-up photographs of the same areas will be taken on Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. |
| Statistical methods | Sample size consideration |
| | Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives. |
| | Data presentations/Descriptive statistics |
| | Three populations will be employed in the analysis of study data. |
| | The intent-to-treat (ITT) population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population. |

- The PK population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters.
- The PD population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the PK and ITT populations, where appropriate.

#### Criteria for evaluation

| Objective | Endpoint |
|---|---|
| Primary | |
| Safety and tolerability of 5 once-<br>weekly IV infusions of SYNT001 to<br>subjects with pemphigus vulgaris or<br>foliaceus | AEs and clinical (safety) laboratory tests |
| Secondary | |
| PK of SYNT001 following a 1-hour IV infusion | PK parameters: $t_{1/2}$ , $C_{max}$ , $T_{max}$ , $AUC_{0\text{-}24}$ , and $AUC_{0\text{-}\infty}$ . |
| Effect of 5 once-weekly IV doses of SYNT001 on: • Total IgG (IgG1-4), IgA, IgM, and albumin • Serum anti-Dsg (1 and 3) antibodies | Changes in levels of IgG, IgG subtypes (IgG1-4), IgA, IgM, albumin, serum anti-Dsg (1 and 3) antibodies |
| Assess immunogenicity | Anti-SYNT001 antibodies |
| Disease Activity | PDAI Scores |
| Exploratory | , |
| Effect of 5 once-weekly IV doses of SYNT001 on biomarkers including: • CIC • C3 • Serum anti-epithelial cell antibody (AECA) levels • Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG) • Immune phenotyping by flow cytometry | Changes in CIC; C3; AECA levels by indirect immunofluorescence; <i>FCGR2A</i> SNP; RNAseq; urine IgG, CD3+CD4+ T, CD3+CD8+ T, monocytes, NK cells and B cells; urine IgG levels; changes in blood transcriptome |
| Concomitant Treatment | Corticosteroid use during the study |
| SYNT001 levels in skin biopsies | Measures of SYNT001 levels in skin biopsies |

Treatment-emergent AEs (TEAEs) will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, or treatment discontinuation will be listed by subject, and cohort using SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken, and outcome.

Laboratory results will be summarized by time point and cohort. The incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the central laboratory. Vital sign measurements will be summarized by cohort at each scheduled time point using descriptive statistics.

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and area under the curve (AUC). PK parameters will be determined using non-compartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

PD results will be summarized by cohort. Descriptive statistics of PD parameters for SYNT001 will include mean, SD, CV, median, minimum, and maximum.

Immunogenicity results will be summarized by cohort. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

**Table 1:** Study Assessments

| | Screening | | | | | | | Tre | atmen | t Perio | d | | | | | | ı | Follow-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepoint (Study Day) | -14 to -1 | 0 | 1<br>(±1<br>hr) | 2<br>(± 2<br>hr) | 5 <sup>p</sup><br>(±4<br>hr) | 7<br>(±6<br>hr) | 12 <sup>p</sup><br>(±6<br>hr) | 14<br>(±6<br>hr) | 19 <sup>p</sup><br>(±6<br>hr) | 21<br>(±6<br>hr) | 28<br>(±6<br>hr) | 29<br>(±1<br>hr) | 30<br>(±2<br>hr) | 33<br>(±4<br>hr) | 42<br>(±3<br>days) | 56<br>(±5<br>days) | 84<br>(±5<br>days) | 112<br>(±5 days) or ET<br>Visit |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Demographics/Medical History | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>a</sup> | X | X | | | | X | | X | | X | X | | | | X | X | X | X |
| Vital Signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse Oximetry <sup>c</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Clinical Safety Labs <sup>d</sup> | X | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | | |
| 12-Lead ECG <sup>f</sup> | X | X | | | | | X | | | | X | | | | | X | | |
| Tetanus & VZV antibodies | | X | | | | | | | | | | | | | | X | X | X |
| PDAI Score | | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| PK Sampling <sup>h</sup> | | X | X | X | X | | | | | | X | X | X | X | | | | |
| Immunogenicity <sup>i</sup> | | X | | | | | | X | | | X | | | | | X | X | X |
| Study Drug Administration <sup>j</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4) <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Xq |
| CIC | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Anti-Dsg (1 & 3) antibody titer | X | X | | | | X | | X | | | | | | X | | X | X | X |
| C3 and AECA <sup>1</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| FCGR2A <sup>m</sup> | | X | | | | | | | | | | | | | | | | |
| RNAseq <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| Urine IgG <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| Immune phenotyping <sup>n</sup> | | X | | | | | | | | | X | | | | | X | | |
| Optional Skin Biopsy | | X | X | X | | | | X | | | | | | X | | X | X | |
| Photography <sup>o</sup> | | X | | | | | | | | | | | | X | | X | X | X |
| Adverse Events | | | | | To be | e collec | ted fron | ı the da | te that t | the ICF | is sign | ed throi | igh the i | ast study | visit | | | |
| Concomitant Medications | | | | | To be | e collec | ted fron | n within | 14 day | s prior | to Day | 0 throu | gh the l | ast study | visit | | | |

ECG = electrocardiogram; ET= Early Termination; HIV = human immunodeficiency virus; ICF = informed consent form; PD = pharmacodynamic; PK = pharmacokinetic; VZV = varicella-zoster virus

Syntimmune, Inc.


Amendment 2.0 Final 12 April 2017


- a: Complete PE, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.
- b: **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. On Days 0, 7, 14, 21, and 28 vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- c: **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d: Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 6.7 for a complete list). Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 112.
- e: **Pregnancy test:** To be performed at time of screening and prior to first dose of SYNT001 on Day 0 and on Days 56 and 112 (urine or serum test is acceptable, however, positive urine tests must be confirmed with serum testing.)
- f: Digital 12-lead ECG to be obtained after 5 minutes of rest in the supine position and in triplicate at least 1-2 minutes apart (see Section 6.6 for additional information). On Days 0 and 28 to be obtained 5 minutes after the completion of infusion. Day 12 ECG will be collected only if the visit is conducted at the study site.
- g: **Serology**: Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 84; if still below the baseline value (or level of detection), the subject will be re-tested at Day 112. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112, will be referred to their primary care physician for further management. See Section 6.7.3 for additional information.
- h: **PK:** Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. See Section 6.7.4 for additional information.
- i: Immunogenicity: Blood samples will be collected pre-dose when collected on dosing days. Samples will be collected on Days 0, 14, 28, 56, 84 and 112. See Section 6.7.6 for additional information.
- j: Prior to **study drug infusion**, SYNT001 drug product is to be diluted in Dextrose 5% in Water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour using a 0.2-micron, inline filter. See Section 9 for additional information.
- k: Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, and IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 6.7.5 for additional information
- 1: Exploratory PD samples (C3 and AECA): collected pre-dose when collected on dosing days. See Section 6.7.5 for complete information.
- m: Samples to be collected and stored; pending review of clinical and pharmacodynamics assessments
- n: Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- o: Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- p: Visit Days 5, 12 and 19 may be conducted via at-home nursing in lieu of a subject visit to the study site.
- q: Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

Table 2: Timing Window Allowances for PK/PD Sampling, ECG, and Vital Sign Measurements

| Pharmacokinetic and Pharmacodynamic Sampling | |
|------------------------------------------------|-------------------------|
| Timepoint | Tolerance Window |
| 0 hour | −240 min to 0 hour |
| 5 minutes post end-of-infusion | ± 5 minutes |
| 2, 4, & 6 hours post end-of-infusion | ± 15 minutes |
| 24 hours post end-of-infusion | $\pm$ 60 minutes |
| 48 hours post end-of-infusion | ± 120 minutes |
| ECG | |
| Timepoint | <b>Tolerance Window</b> |
| 5 minutes post end-of-infusion | ± 10 minutes |
| Vital Signs <sup>a</sup> | |
| Timepoint | <b>Tolerance Window</b> |
| 0 hour | −240 min to 0 hour |
| 15, 30, and 45 minutes after start of infusion | ± 5 minutes |
| 60 minutes after start of infusion | ± 10 minutes |
| 30, 60 and 120 minutes post end-of-infusion | ± 10 minutes |

a. Vital signs to include blood pressure, pulse rate, respiratory rate, oral temperature, and pulse oximetry.

## TABLE OF CONTENTS

| PROCE | EDURES IN CASE OF EMERGENCY | 3 |
|--------|---------------------------------------------|----|
| INVEST | TIGATOR SIGNATURE | 4 |
| 1 SY | YNOPSIS | 5 |
| LIST O | F ABBREVIATIONS | 24 |
| 2 B | ACKGROUND AND RATIONALE | 26 |
| 2.1 | Study Rationale | 27 |
| 2.2 | Selection of Doses in this Study | |
| 2.3 | Compliance Statement | |
| 3 S7 | TUDY OBJECTIVES | 29 |
| 3.1 | Primary Objective | 29 |
| 3.2 | Secondary Objectives | 29 |
| 3.3 | Exploratory Objectives | 29 |
| 4 S7 | TUDY DESIGN | 30 |
| 4.1 | Study Sites | 30 |
| 4.2 | Study Endpoints | 30 |
| 4.3 | Overview of Study Design | 31 |
| 4.4 | Randomization and Blinding | 33 |
| 5 S7 | TUDY POPULATION | 34 |
| 5.1 | Target Population | 34 |
| 5.2 | Inclusion Criteria | 34 |
| 5.3 | Exclusion Criteria | 35 |
| 6 S7 | TUDY PROCEDURES | 37 |
| 6.1 | Informed Consent | 37 |
| 6.2 | Demographics and Medical History | 37 |
| 6.3 | | |
| 6.4 | Pemphigus Disease Area Index (PDAI) Scoring | 37 |
| 6.5 | Vital Sign Measurements | 37 |
| 6.6 | 12-Lead Electrocardiogram (ECG) | |
| 6.7 | Clinical Laboratory Measurements | |
| | 6.7.1 Pregnancy Testing | |
| | 6.7.2 Virology | 40 |

| | | 6.7.3 | Serum Tetanus Antibody and Varicella-Zoster Virus Antibody | dy Testing40 |
|---|---|---|---|---|
| | | 6.7.4 | Pharmacokinetics (PK) Sampling | 40 |
| | | 6.7.5 | Pharmacodynamic Sampling | 41 |
| | | 6.7.6 | Immunogenicity Testing | 42 |
| | 6.8 | Study | y Drug Administration | 43 |
| | 6.9 | Prior | and Concomitant Medications | 43 |
| | 6.10 | Adve | erse Event Assessments | 43 |
| | 6.11 | Photo | ographs | 44 |
| | 6.12 | Skin | Biopsy | 44 |
| 7 | ST | UDY A | SSESSMENTS | 45 |
| | 7.1 | Scree | ening Period: Day -14 to Day -1 | 45 |
| | 7.2 | | Ilment and First Treatment: Day 0 | |
| | 7.3 | Follo | w-up: Day 1 | 47 |
| | 7.4 | Follow-up: Day 2 | | |
| | 7.5 | Follo | w-up: Day 5 | 48 |
| | 7.6 | Treat | ment Day 7 (Dose 2) | 48 |
| | 7.7 | Dose | 2 Follow-up Day 12 | 49 |
| | 7.8 | Treat | ment Day 14 (Dose 3) | 49 |
| | 7.9 | Dose | 3 Follow-up Day 19 | 51 |
| | 7.10 | Treat | ment Day 21 (Dose 4) | 51 |
| | 7.11 | Treat | ment Day 28 (Dose 5) | 52 |
| | 7.12 | Follo | w-up Day 29 | 53 |
| | 7.13 | Follo | w-up Day 30 | 54 |
| | 7.14 | Follo | w-up Day 33 | 54 |
| | 7.15 | Follo | w-up Day 42 | 55 |
| | 7.16 | Follo | w-up Day 56 | 55 |
| | 7.17 | Follo | w-up Day 84 | 56 |
| | 7.18 | Follo | w-up Day 112 (End-of-Study) or Early Termination Visit | 57 |
| 8 | RE | MOVIN | NG SUBJECTS FROM STUDY | 58 |
| | 8.1 | Subje | ect Withdrawal | 58 |
| | 8.2 | Study Discontinuation | | |
| | 8.3 | Repla | acements | 59 |
| | 8.4 | Stopp | ping Rule | 59 |
| | | 8.4.1 | Dose-Escalation Stopping Rule | 59 |
| | | 8.4.2 | Study Stopping Rule | 60 |
| | | 8.4.3 | Individual Stopping Rule | 60 |

| 9 | ST | UDY DR | UG | 61 |
|---|---|---|---|---|
| | 9.1 | SYNT | 001 | 61 |
| | 9.2 | Cohor | t Dosing | 61 |
| | 9.3 | | g of Dosing | |
| | 9.4 | | y of Investigational Products | |
| | 9.5 | | gational Product Retention at Study Site | |
| | 9.6 | | ngs and Precautions | |
| | | 9.6.1 | Infusion Reaction | |
| | | 9.6.2 | Potential Immune Effects | 67 |
| 10 | CC | NCOMI | ΓΑΝΤ MEDICATION AND TREATMENT | 69 |
| 11 | SA | FETY | | 71 |
| | 11.1 | Safety | Parameters | 71 |
| | 11.2 | Advers | se Event Definition | 71 |
| | 11.3 | Evalua | ting Adverse Events | 72 |
| | | 11.3.1 | Serious Adverse Events | 72 |
| | | 11.3.2 | Overdose | 73 |
| | | 11.3.3 | Non-Serious Adverse Events | 73 |
| | | 11.3.4 | Protocol-Related Adverse Events | 73 |
| | | 11.3.5 | Assessment of Causality | 73 |
| | | 11.3.6 | Recording Adverse Events | 74 |
| | | 11.3.7 | Planned Hospitalization | 74 |
| | | 11.3.8 | Reporting Pregnancies | 75 |
| | | 11.3.9 | Serious Adverse Event Reporting | 75 |
| | | 11.3.9.1 | Governing Regulatory Requirements | 75 |
| | | 11.3.9.2 | Time Frame for Reporting | 76 |
| | | 11.3.9.3 | Information to be Provided by the Investigator | 77 |
| | | 11.3.10 | Regulatory Reporting | 78 |
| | | 11.3.11 | Follow-up Information on a Serious Adverse Event (SAE) | 79 |
| | 11.4 | Other | Safety Considerations | 79 |
| | | 11.4.1 | Laboratory Data | 79 |
| | | 11.4.2 | Medication Errors | 79 |
| | | 11.4.3 | Follow-Up of Adverse Events | 79 |
| | 11.5 | Safety | Monitoring for Dose Escalation | 79 |
| 12 | ST | ATISTIC | AL CONSIDERATIONS | 81 |
| | 12.1 | Genera | al Design | 81 |
| | 12.2 | | e Size Justification | |
| | 12.3 | Statist | ical Considerations | 81 |

| | | 12.3.1 | Study Populations | 81 |
|---|---|---|---|---|
| | | 12.3.2 | Subject Accountability, Demographics, and Baseline Character | ristics 82 |
| | | 12.3.3 | Concomitant Medications | 82 |
| | 12.4 | Plann | ed PK Analysis | 82 |
| | 12.5 | Safety | Data | 83 |
| | 12.6 | | nacodynamic/Activity Data | |
| | 12.7 | Immu | nogenicity Data | 83 |
| | 12.8 | Interin | n Analysis | 84 |
| 13 | DA | ATA QU | ALITY ASSURANCE | 85 |
| 14 | ST | UDY AI | OMINISTRATION | 86 |
| | 14.1 | Study | Administrative Structure | 86 |
| | 14.2 | Ethica | al Conduct of the Study | 86 |
| | 14.3 | Inforn | ned Consent (ICF) | 86 |
| | 14.4 | Institu | ntional Review Board | 87 |
| | 14.5 | Dose | Escalation Committee | 87 |
| | 14.6 | Future | e Use of Subject Samples | 88 |
| 15 | CC | ONDITIC | ONS FOR MODIFYING THE PROTOCOL | 89 |
| 16 | CC | ONDITIC | ONS FOR TERMINATING THE STUDY | 90 |
| 17 | ST | UDY DO | OCUMENTATION, CRFS, AND RECORD KEEPING | 91 |
| | 17.1 | Invest | igator's Files and Retention of Documents | 91 |
| | 17.2 | Sourc | e Documents and Background Data | 91 |
| | 17.3 | Audit | s and Inspections | 92 |
| | 17.4 | Electr | onic Case Report Forms | 93 |
| 18 | Mo | ONITOR | ING THE STUDY | 94 |
| 19 | CC | ONFIDEN | NTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECOR | RDS95 |
| 20 | PU | BLICAT | TION OF DATA AND PROTECTION OF TRADE SECRETS | 96 |
| 21 | DE | EEDENI | OEC. | 07 |

| LIST | <b>OF</b> | TA | BI | ES |
|------|-----------|----|----|----|
|------|-----------|----|----|----|

| Table 1: | Study Assessments | 16 |
|---|---|---|
| Table 2: | Timing Window Allowances for PK/PD Sampling, ECG, and Vital Sig | gn |
| | Measurements | 18 |
| Table 3: | Clinical Laboratory Panels | 39 |
| Table 4: | Pharmacodynamic/ Activity Assessments | 42 |
| Table 5: | Grading and Management of Allergic or Infusion-Related Reactions | 66 |
| Table 6: | Study Administrative Structure | 86 |
| _ | Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions | |
| _ | Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions Management of Severe (Grade 3 or higher) Infusion Reactions | |
| LICE OF | | |
| | APPENDICES | |
| Appendix A | A: NCI CTCAE, Version 4.03 | 99 |
| Appendix F | 3: Pemphigus Disease Area Index | 100 |

### LIST OF ABBREVIATIONS

ADA Anti-drug antibodies

AE Adverse event

AECA Anti-epithelial cell antibody
ALT Alanine aminotransferase
ANA Antinuclear antibody
AST Aspartate aminotransferase
ATC Anatomical therapeutic chemical

AUC<sub>0-24</sub> Area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose

 $AUC_{0-\infty}$  Area under the plasma concentration-time curve from pre-dose (time 0) to infinity

BLQ Below the limit of quantification

BMI Body mass index
BUN Blood urea nitrogen

CAR-T Chimeric antigen receptor and T-cell

CFR Code of Federal Regulations
C3 Complement component 3
CBC Complete blood count

CIC Circulating immune complexes

CIDP Chronic inflammatory demyelinating polyneuropathy

C<sub>max</sub> Maximum plasma concentration determined directly from the concentration-time profile

CRO Contract research organization

CV Coefficient of variation

CVID Common variable immune deficiency

DEC Dose escalation committee
D5W Dextrose 5% in Water
DIF Direct immunofluorescence
DNA Deoxyribonucleic acid
ECG Electrocardiogram

eCRF Electronic case report form
ESR Erythrocyte sedimentation rate
FcGR2a Fc Gamma R2a receptor
FcRn Neonatal Fc receptor

FDA Food and Drug Administration

GCP Good Clinical Practice

GI Gastrointestinal
HBV Hepatitis B virus
HCV Hepatitis C virus

HIPAA Health Insurance Portability and Accountability Act

HIV Human immunodeficiency virus

IB Investigator's brochure IC Immune complex

ICF Informed consent form

ICH International Conference on Harmonization

IgA Immunoglobulin A
IgG Immunoglobulin G
IgG1-4 Immunoglobulin G1-G4
IgM Immunoglobulin M
IL-12 Interleukin 12

IND Investigational new drug
IRB Institutional review board

ITT Intent-to-treat
IUD Intrauterine devices

IV Intravenous

IVIG Intravenous immunoglobulin

MedDRA Medical Dictionary for Regulatory Activities

NHL Non-Hodgkin lymphoma
PD Pharmacodynamics
PE Physical examination
PK Pharmacokinetic
RBC Red blood cells
RNAseq RNA sequencing

QTcF Corrected QT interval using Fridericia's formula

SAE Serious adverse event
SAP Statistical analysis plan
SAS Statistical Analysis System

SD Standard deviation

SNP Single nucleotide polymorphism

SOC System Organ Class

SOP Standard operating procedures

SYNT001 A humanized, affinity matured IgG4-kappa monoclonal antibody

 $t_{1/2}$  Half-life

TEAE Treatment-emergent adverse event

T<sub>max</sub> Observed time to reach peak plasma concentration

TNF Tumor necrosis factor ULN Upper limit of normal

UNS Unscheduled

VZV Varicella-zoster virus

WAIHA Warm antibody autoimmune hemolytic anemia

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

### 2 BACKGROUND AND RATIONALE

SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG ICs from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG-containing ICs further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen-presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG ICs within and among compartments important in cellular immunity, it is anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8<sup>+</sup> and CD4<sup>+</sup> T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG that are involved in certain autoimmune conditions and dismantle their ability to cause disease.

SYNT001 targets key mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP).

While current treatments for certain autoimmune disorders, including high-dose steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are associated with significant adverse effects, as well as delayed or non-durable responses.

Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies have been shown to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, which significantly decreases total IgG, including a corresponding decrease in the level of the pathogenic autoantibodies and the ICs to which they are associated, may lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification.

### 2.1 Study Rationale

This study is being conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers.

### 2.2 Selection of Doses in this Study

The planned dose levels of SYNT001 for this Phase 1b safety and proof-of-concept study of 10 mg/kg and 30 mg/kg were selected from careful review of the safety, tolerability, and PD effect on total IgG levels after single and repeat dosing of SYNT001 in non-human primates (NHPs), as well as the safety, tolerability, and PD effect on total IgG levels after single ascending doses of SYNT001 in healthy volunteers. In addition, further consideration was given to the desired level of FcRn blockade to achieve suppression of IgG to a range that has been previously correlated with disease remission. Further, we considered the potential effects of inhibiting FcRn function as they relate to immune complex associated innate and adaptive immunity in choosing these dose levels based upon exploratory studies of a single ascending dose of SYNT001 in healthy volunteers. From the NHP studies, single doses of SYNT001 produced a dose-dependent decrease in total IgG and a further decrease was seen with repeated weekly doses up to a maximum 70% reduction at 100 mg/kg. This magnitude of total IgG reduction is approaching the expected maximal effect of 100% inhibition of FcRn function based on murine studies also performed by Syntimmune and others [Roopenian 2003, Nixon 2015]. In the recently completed Phase 1a trial with SYNT001 in healthy volunteers a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the NHP studies further reductions are expected following multiple dosing. A comparable decrease in pathogenic autoantibodies is also anticipated.

In the NHP studies, relevant adverse effects, mild-to-moderate infusion reactions, were observed only after the third weekly IV administration, concurrent with the development of anti-SYNT001 antibodies. In the recently completed Phase 1a healthy male volunteer study, the doses of SYNT001 up to and including 30 mg/kg have been well tolerated. There were no dose limiting toxicities, serious adverse events, or any other safety concerns identified. No AEs were observed in the 1 and 3 mg/kg dose cohorts. A single Grade 2 AE was observed; a headache in the 10 mg/kg cohort, treated with acetaminophen. Other subjects had mild (Grade 1) AEs at 10 mg/kg. In Cohort 4 (30 mg/kg), 5 subjects received SYNT001. All five subjects experienced AEs; all were mild (Grade 1), transient and resolved spontaneously without intervention. Therefore, it is anticipated that the doses selected for this study should be well tolerated and have clinically relevant PD effects in patients with chronic pemphigus (vulgaris or foliaceus). For a summary of

findings from the single dose, clinical study in healthy subjects and further details on the nonclinical findings, please refer to the SYNT001 Investigator's Brochure.

# 2.3 Compliance Statement

This study will be conducted in compliance with Good Clinical Practice (GCP), including the International Conference on Harmonisation (ICH) Guidelines and FDA regulations, consistent with the principles outlined in the Declaration of Helsinki. In addition, the Investigator agrees to adhere to all applicable local laws and regulatory requirements relevant to the use of new therapeutic agents.

The study will be conducted in compliance with the protocol. The appropriate Institutional Review Boards (IRBs) must approve the protocol, any amendments, and the subject informed consent form (ICF) prior to implementation.

Freely given written informed consent must be obtained from every subject prior to participation in this clinical trial. As part of this procedure, the Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or AEs that may occur. The study subject should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The Investigator or designee will provide the Sponsor with a copy of the IRB-approved informed consent form prior to the start of the study. The rights, safety, and well-being of participating subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (e.g., loss of medical licensure, debarment).

#### 3 STUDY OBJECTIVES

### 3.1 Primary Objective

The primary objective of this study is to evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus).

### 3.2 Secondary Objectives

The secondary objectives of this study are as follow:

- To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers:
  - o Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM
  - o Albumin
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers:
  - o Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
  - o Pemphigus Disease Area Index (PDAI)
- To assess immunogenicity (anti-SYNT001 antibodies)

### 3.3 Exploratory Objectives

The exploratory objectives of this study are as follow:

- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including:
  - o Serum anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence
  - o Circulating immune complexes (CIC)
  - o Complement component 3 (C3)
  - Exploratory biomarkers (FCGR2A single nucleotide polymorphism-SNP, RNAseq, urine IgG)
  - Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
  - o SYNT001 levels in skin biopsies (optional)
- To characterize corticosteroid use during the study

#### 4 STUDY DESIGN

## 4.1 Study Sites

This study will be conducted at approximately 10 sites in the United States (US).

### 4.2 Study Endpoints

**Primary Outcome Measures:** Assessment of safety data (adverse events [AEs], serious adverse events [SAEs], vital sign measurements, ECGs and clinical laboratory tests) will be the primary safety measure.

### **Secondary Outcome Measures**

#### Pharmacokinetics:

Half-life (t<sub>1/2</sub>), maximum plasma concentration determined directly from the
concentration-time profile (C<sub>max</sub>), observed time to reach peak plasma concentration
(T<sub>max</sub>), area under the plasma concentration-time curve from pre-dose (time 0) to
24 hours post-dose (AUC<sub>0-24</sub>), and area under the plasma concentration-time curve
from pre-dose (time 0) to infinity (AUC<sub>0-∞</sub>)

### PD Biomarkers:

- Ig Assessments: Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o IgA levels
  - o IgM levels
- Albumin levels

### Disease activity markers:

- Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
- Pemphigus Disease Area Index (PDAI) scores

### Immunogenicity:

• Anti-SYNT001 antibodies

### **Exploratory Outcome Measures**

Biomarkers, including:

- CIC
- C3
- Serum AECA levels
- Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG)

- Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- SYNT001 levels in skin biopsies (optional)

#### **Concomitant Treatments**

Corticosteroid use

Further details on the statistical and analytical plan for these endpoints are available in Section 12, Statistical Considerations.

### 4.3 Overview of Study Design

This will be a multicenter, open-label study to assess the safety, tolerability, activity, PK, PD, and immunogenicity of 5 once-weekly IV infusions of SYNT001 to subjects with chronic pemphigus (vulgaris or foliaceus).

Planned doses of SYNT001 to be studied are 10 mg/kg and up to 30 mg/kg. Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 10 mg/kg or up to 30 mg/kg. Based on review of safety, PD, and clinical outcomes of the first cohort, the dose for the second cohort may be adjusted, but with a maximum dose of 30 mg/kg. Based on review of safety, PD and clinical outcomes from these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of<br>Subjects | Dose |
|--------|--------------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All data through Day 42

(2 weeks after the last subject's last dose in Cohort 1) will be reviewed before Cohort 2 is initiated. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule.

Safety evaluations will be conducted by a dose escalation committee (DEC). The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions. Dosing and dose escalation will proceed if the DEC has determined that it would be safe and appropriate to do so. In addition, over the course of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84, and 112. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42 and 56 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects also will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, AE assessments, concomitant medication assessments, and electrocardiograms (ECG).

**Note**: No vaccinations may be given from within 2 weeks of screening through Day 56. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator.

# 4.4 Randomization and Blinding

This is an open-label study.

#### 5 STUDY POPULATION

### 5.1 Target Population

This study will be conducted in approximately 16 male and female subjects (2 cohorts of 8 subjects each) with a confirmed diagnosis of pemphigus (vulgaris or foliaceus); however, a third cohort of up to 8 subjects may be added. Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled visits. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects may be enrolled with pemphigus foliaceus.

#### 5.2 Inclusion Criteria

A subject must meet the following criteria to be eligible for the study:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq$  18 years of age;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal;
  - c. History of at least one positive tissue based test (biopsy, DIF)
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose > 12 months prior to screening;
  - b. If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
  - c. If being treated with corticosteroids, must be ≤ 1mg/kg/day and stable (< 10% change in dose) for 2 weeks prior to screening;

- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 35.0 \text{ kg/m}^2$ ;
- 6. Has a negative urine pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through the final study visit.

### 5.3 Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

- 1. Unable or unwilling to comply with the protocol;
- Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG treatment within 60 days of screening;
- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;

- 8. Any exposure to an investigational drug or device within 30 days prior to screening;
- 9. Plasmapheresis or immunoadsorption within 60 days of screening
- 10. Cellular therapy at any time prior to screening
- 11. Use of any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of screening;
- 12. Serum total IgG < 600 mg/dL;
- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (e.g., a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results);
- 14. Any vaccination within 2 weeks of screening

#### 6 STUDY PROCEDURES

#### 6.1 Informed Consent

All subjects must take part in the informed consent process. Adequate time must be allowed for the subject to ask questions and make a voluntary decision. No protocol-specific procedures, including screening procedures, are to be performed until the subject has signed and dated an IRB-approved ICF. Subjects may withdraw consent at any time. Participation in the study may be terminated at any time without the subject's consent as determined by the Investigator.

# **6.2** Demographics and Medical History

Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and eCRF. Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery and concomitant treatments.

### 6.3 Physical Examination

A complete physical examination will be performed as outlined in Table 1. The complete PE will include measurements of weight (in kg) and height (in cm; height to be measured only at screening visit) and a review of the following body systems:

- General appearance
- Head, eyes, ears, nose, and throat
- Neck
- Respiratory
- Cardiovascular
- Abdomen
- Neurologic
- Extremities
- Dermatologic
- Lymphatic

Any abnormal and clinically significant findings from the PE must be recorded in the appropriate eCRF. Findings at screening and Day 0 (pre-dose) will be recorded as medical history.

### 6.4 Pemphigus Disease Area Index (PDAI) Scoring

Pemphigus severity and disease activity will be measured using the PDAI. See Appendix B.

### 6.5 Vital Sign Measurements

Vital sign measurements will be collected after the subject has been sitting for 5 minutes. Vital sign assessments will include measurements of sitting blood pressure (mm Hg), heart rate (beats

per minute), respiration rate (breaths per minute), oral temperature (Celsius). Abnormal results are to be repeated after 5 minutes of rest. Pulse oximetry (%) also is to be measured. See Table 2 for timing window allowances with respect to measurement collection.

On Days 0, 7, 14, 21, and 28, vital sign measurements are to be obtained immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion. Details on the management of mild to moderate and severe infusion reactions can be found in Figure 1 and Figure 2. Abnormalities in vital sign measurements will be graded in severity per the NCI CTCAE scale Version 4.03.

Subjects should be seated quietly for at least 5 minutes in a chair with their backs supported, their feet flat on floor (legs uncrossed), and their arms bared on a hard surface, with the arm slightly abducted and bent, with palm up and the midpoint of upper arm at heart level. Correct cuff and bladder size should be utilized and the same cuff and arm should be used per subject throughout study.

### 6.6 12-Lead Electrocardiogram (ECG)

Digital 12-lead ECG measurements will be obtained at screening, on Days 0 and 28 at 5 minutes after the completion of the infusion and at the Day 56 visit. Subjects who conduct their Day 12 visit at the investigative site, as opposed to an at-home nurse visit, will have an additional ECG performed. ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each 1 to 2 minutes apart. See Table 2 for timing window allowances with respect to performing ECG.

The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant.

Normal QTcF is  $\leq 450$  msec.

Abnormalities in the ECG that appear following therapy or that result in clinical signs and symptoms are considered clinically significant for the purposes of this study and will be recorded on the AE eCRF.

### 6.7 Clinical Laboratory Measurements

Collection time for all safety, PD, and exploratory labs are outlined in Table 1.

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and anti-drug antibody samples) will be performed using established methods by a central laboratory. Safety laboratory panels are defined as listed in Table 3. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and anti-drug antibody samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 112. The total blood draw for each subject who completes the study at Day 112, will be approximately 381 mL. Please refer to the Laboratory Manual for more information.

**Table 3: Clinical Laboratory Panels** 

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| CBC with differential and blood smear Erythrocyte Sedimentation Rate (ESR) | <ul> <li>Albumin</li> <li>Alkaline phosphatase</li> <li>ALT</li> <li>AST</li> <li>BUN</li> <li>Calcium</li> <li>Carbon dioxide</li> <li>Chloride</li> <li>Creatinine</li> <li>Glucose</li> <li>LDH</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total and direct bilirubin</li> <li>Total protein</li> <li>Uric acid</li> <li>C-Reactive Protein</li> </ul> | <ul> <li>Appearance</li> <li>Color</li> <li>pH</li> <li>Specific gravity</li> <li>Ketones</li> <li>Protein</li> <li>Glucose</li> <li>Nitrite</li> <li>Urobilinogen</li> <li>Blood/hemoglobin</li> <li>Leukocyte esterase</li> <li>Bilirubin</li> <li>Microscopic examination of sediment: only if the results of the urinalysis dipstick evaluation are positive for blood/hemoglobin</li> </ul> |
| Virology | | |
| <ul><li>Hepatitis C</li><li>Hepatitis B</li></ul> | | |

- HIV
- VZV
- Tetanus

ALT = alanine aminotransferase; AST = aspartate aminotransferase; CBC = complete blood count; BUN = blood urea nitrogen; HIV = human immunodeficiency virus; LDH = lactate dehydrogenase; VZV = varicella-zoster virus

Abnormalities in clinical laboratory tests that are considered clinically significant are to be recorded on the AE electronic case report form (eCRF) page. Laboratory results will be graded using the NCI CTCAE, Version 4.03. If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as an SAE (see Section 11.3.1).

### 6.7.1 Pregnancy Testing

Pregnancy testing will be performed for women of childbearing potential at screening and prior to first dose of SYNT001 on Day 0 and Days 56 and 112 (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing.)

### 6.7.2 Virology

Testing for HCV antibody, hepatitis B surface antigen, and HIV antibody will be performed at screening.

### 6.7.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

Samples for serum tetanus antibody and varicella-zoster virus antibody testing are to be collected at baseline (pre-dose, Day 0) and on Day 56 (Follow-Up visit). Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. Specifically, if the baseline VZV titer is above the detectable level, but tetanus is not, only the VZV antibody titer will be tested on Day 56. If the Day 56 results are below the baseline value, defined as greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 84; if still below the baseline value (or level of detection), the subject will be re-tested at Day 112. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112, will be referred to their primary care physician for further management.

### 6.7.4 Pharmacokinetics (PK) Sampling

Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug

infusion. Additional samples will be collected on Days 5 and 33. The actual time and date of each blood draw is to be recorded.

Study drug concentration will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-24}$ , and  $AUC_{0-\infty}$ .

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual

### 6.7.5 Pharmacodynamic Sampling

PD samples will be collected for analyses throughout the study. On Days 0, 7, 14, 21, and 28, samples should be collected prior to infusion of study drug. Measurements for albumin PD biomarkers will be derived from the clinical safety laboratory results. Samples for each type of PD will be collected according to the schedule shown in **Table 4**.

Table 4: Pharmacodynamic/ Activity Assessments

| Parameter | Collection Timepoints |
|---|---|
| IgG, IgG subtypes (IgG1-4), IgA, IgM | Screening, and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, 56, 84 and 112. |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84 and 112 |
| • Albumin | Screening, and Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 112 |
| Anti-Dsg (1 and 3) antibody titer | Screening, Days 0, 7, 14, 33, 56, 84 and 112 |
| <ul> <li>Complement component 3 (C3)</li> <li>Anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence</li> </ul> | Days 0, 14, 33, 56, 84 and 112 |
| Exploratory biomarker (RNAseq, Urine IgG) | Days 0, 14, 33, 56, 84 and 112 |
| Immune phenotyping by flow cytometry for<br>measurement of CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T,<br>monocytes, NK cells and B cells | Days 0, 28 and 56 |
| Exploratory biomarker (FCGR2A SNP) | Day 0 |

See Table 2 for timing window allowances with respect to measurement collection. Detailed instructions for sample collection (including collection tubes) and preparation will be provided in a separate laboratory manual.

### 6.7.6 Immunogenicity Testing

Serum samples will be collected for immunogenicity analyses on Days 0 (pre-dose), 14, 28, 56, 84 and 112.

SYNT001 is being developed for the acute and chronic therapy of autoimmune disorders. Although SYNT001 is a humanized IgG4 monoclonal antibody, exposure to SYNT001 in clinical trials could result in the development of anti-drug antibodies (ADAs), with potential consequences ranging from neutralization or lessening of drug efficacy to safety consequences such as allergic reactions. Testing will first detect binding ADAs, then, for all confirmed positive samples, there will be testing for neutralizing effects.

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

#### 6.8 **Study Drug Administration**

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute IV infusions of SYNT001 10 mg/kg or up to 30 mg/kg. SYNT001 will be given as a 250-mL IV infusion over 1 hour using a 0.2-micron, inline filter. Based on review of safety data, as well as available and relevant PD results, and clinical outcomes of Cohort 1, a decision about proceeding with Cohort 2 will be made. Based on review of all safety data, available PD results, and clinical outcomes of these 2 cohorts, a third cohort of 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort No. | Study Drug | Dose Level<br>(mg/kg/dose) |
|------------|------------|----------------------------|
| 1 | SYNT001 | 10 mg/kg |
| 2 | SYNT001 | 30 mg/kg |

See Section 9.1 for dosing schedule.

#### 6.9 **Prior and Concomitant Medications**

All medications a subject receives within 14 days prior to enrollment through the end of the study will be documented on the source document and eCRF.

Note: No vaccinations may be given from within 2 weeks of screening through Day 56. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator.

#### 6.10 **Adverse Event Assessments**

Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form and continuing through the last study visit. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE.

Clinical AEs will be graded using the NCI CTCAE, Version 4.03 (Appendix A).

**Note:** AEs resulting in a subject's permanent discontinuation from the study, regardless of seriousness or relationship to study drug, MUST be promptly reported to the sponsor. Additionally, subjects must be followed until return to normal and/or resolution of the AE.

See Section 11 for more information.

### 6.11 Photographs

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

## 6.12 Skin Biopsy

Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33, 56 and 84 to analyze SYNT001 levels.

### 7 STUDY ASSESSMENTS

### 7.1 Screening Period: Day -14 to Day -1

Informed consent must be obtained before any study-specific samples are taken or study-specific tests or evaluations are conducted. The following assessments at the screening visit are to occur within 14 days before dosing. Study eligibility will be based on satisfying all the study inclusion and exclusion criteria.

At the screening visit, information will be collected and subjects will have clinical evaluations as follows:

- Informed consent (Section 6.1)
- Medical history and demographic data (Section 6.2)
- Review inclusion and exclusion criteria (Section 5.2, Section 5.3)
- Complete PE, including height and weight (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Section 6.6)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Hepatitis and HIV screen (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.2 Enrollment and First Treatment: Day 0

Study Day 0 is defined as the date the subject is administered their first dose of study drug. On Day 0, subjects will be asked to come to the clinic and the following procedures will be performed prior to the first dose of study drug:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody (Section 6.7)
- PDAI Score (Section 6.4)
- PK baseline sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - FCGR2A SNP
  - RNAseq
  - Urine IgG
  - Immune phenotyping
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral

temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)

- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.3 Follow-up: Day 1

On Day 1 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.4 Follow-up: Day 2

On Day 2 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.5 Follow-up: Day 5

On Day 5 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 0), subjects may return to the clinic or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.6 Treatment Day 7 (Dose 2)

On Day 7 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion

Protocol SYNT001-103

and at completion of the infusion (Section 6.5)

- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.7 Dose 2 Follow-up Day 12

On Day 12 ( $\pm$  6 hours) the subject may return to the clinic, or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
- If visit performed at the study site: 12-Lead ECG to be obtained in triplicate (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.8 Treatment Day 14 (Dose 3)

On Day 14 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)

- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.9 Dose 3 Follow-up Day 19

On Day 19 (± 6 hours) the subject may return to the clinic, or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.10 **Treatment Day 21 (Dose 4)**

On Day 21,  $(\pm 6 \text{ hours})$  subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)

• AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.11 Treatment Day 28 (Dose 5)

On Day 28 ( $\pm$  6 hours), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (collected just prior to the start of the study drug infusion; record collection date and time for each PK sample) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Immune phenotyping
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion

- and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.12 Follow-up Day 29

On Day 29 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.13 Follow-up Day 30

On Day 30 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.14 Follow-up Day 33

On Day 33 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 28), subjects will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

Protocol SYNT001-103

#### 7.15 Follow-up Day 42

On Day 42 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.16 Follow-up Day 56

On Day 56 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section
- Pregnancy test (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the sitting position) (Section 6.6)
- Serum tetanus antibody and VZV antibody; Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer

- C3
- AECA
- RNAseq
- Urine IgG
- Immune phenotyping
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.17 Follow-up Day 84

On Day 84 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Serum tetanus antibody and VZV antibody testing if required. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

Protocol SYNT001-103

# 7.18 Follow-up Day 112 (End-of-Study) or Early Termination Visit

On Day 112 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody testing if required. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 8 REMOVING SUBJECTS FROM STUDY

Every reasonable effort will be made to keep the subject in the study; however, if a subject is withdrawn from the study, every effort will be made by the Investigator to complete and report the reasons for withdrawal as thoroughly as possible. The reason(s) for termination must be clearly documented on the appropriate page of the eCRF. Once a subject discontinues from the study for any reason, every effort will be made to collect all clinical and laboratory data as scheduled for the Early Termination Visit (See Table 1). A termination eCRF must be completed for all enrolled subjects.

# 8.1 Subject Withdrawal

A subject's participation in the study may be prematurely discontinued for any of the following reasons:

- 1. The subject wishes to withdraw from the study.
- 2. Request by a regulatory agency (e.g., Institutional Review Board).
- 3. Subject experiences a significant or intolerable AE.
- 4. The subject experiences a significant adverse change in vital signs, PE findings, or a clinical laboratory parameter.
- 5. The subject has a need for a concomitant medication that is not permitted by the study protocol.
- 6. The subject experiences generalized impairment or mental incompetence that would result in the subject being unable to understand his or her participation in the study.
- 7. If, in the Investigator's medical judgment, further participation would be injurious to the health and well-being of the subject, or is not in the best interest of the subject.
- 8. Administrative reasons, such as subject non-compliance or a major protocol violation.

Subjects who are withdrawn from this study due to an AE determined to be related to study drug are to be followed until there is either:

- Resolution or stabilization of the AE determined to be related
- The subject is lost to follow-up
- The event is otherwise explained

If there is a persistent AE contributing to discontinuation that is determined to be related to SYNT001, subjects must be followed with appropriate medical management until resolution or stabilization.

A reasonable effort should be made to contact any subject lost to follow-up during the study to complete assessments and retrieve any outstanding data. If the subjects are unreachable by telephone after three (3) attempts, the minimum of a registered letter should be sent requesting that contact be made with the Investigator to report survival information.

### 8.2 Study Discontinuation

Syntimmune Inc. has the right to terminate or to stop the study at any time. Reasons for study discontinuation may include, but are not limited to the following:

- The incidence or severity of AEs in this or other related studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Drug supply issues
- Excessive subject self-withdrawal
- Significant protocol violations (e.g., violation of eligibility criteria, dosing errors, missing data for study endpoint analysis)

## 8.3 Replacements

Enrolled subjects withdrawn for a reason other than an AE will be replaced if they have not been dosed or have only received one dose of study drug at the time of discontinuation, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled study visits.

# 8.4 Stopping Rule

## 8.4.1 Dose-Escalation Stopping Rule

Dose escalation decisions will be made by a Dose Escalation Committee (DEC) and will be based on safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities, AEs, SAEs, and total IgG levels.

Dose-limiting toxicity (DLT) will be defined generally as severe (Grade 3) AEs occurring in  $\geq$ 2 subjects that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. If the dose-escalation stopping rule is met during Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics will be reviewed and the cohort may resume (if applicable) or a new cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met in Cohort 1, dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met for the first time during Cohort 2, all safety data and all available pharmacodynamics will be reviewed and the cohort may resume (if applicable) or a new cohort may be added at a dose a minimum of 30% lower than the Cohort 2 dose. If the stopping rule is not met in Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data.

## 8.4.2 Study Stopping Rule

If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects.

### 8.4.3 Individual Stopping Rule

Dosing for any individual subject will be discontinued (i.e., no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject will be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus.

### 9 STUDY DRUG

For detailed information regarding SYNT001 preparation and administration, refer to the Pharmacy Manual.

### 9.1 SYNT001

SYNT001 is provided in vials containing 5 mL SYNT001 (extractable volume) at a nominal concentration of 50 mg/mL. The product is supplied as a liquid at pH  $6.5 \pm 0.5$ . SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for infusion. SYNT001 will be infused via IV in 250 mL over 1 hour using a 0.2-micron, inline filter.

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these two cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

The specification for host cell DNA in SYNT001 is < 2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing is limited to 5000 mg of SYNT001. Therefore, at the highest dose possible in this study (45 mg/kg), maximum subject weight will be limited to 111 kg.

## 9.2 Cohort Dosing

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. Cohort 2, and Cohort 3 if added, will be dosed per the same schedule

### 9.3 Timing of Dosing

On Days 0, 7, 14, 21, and 28, subjects will receive a 60-minute IV infusion of SYNT001 in the morning. The date and time the dose is administered will be recorded.

### 9.4 Identity of Investigational Products

All supplies of SYNT001 will be supplied by Syntimmune and must be stored refrigerated (2°C to 8°C/36°F to 46°F) in the carton and protected from light, in a securely locked area, accessible to authorized persons only, until needed for dose preparation. Qualified site personnel will

inventory the investigational product received and will maintain records of disposition of the drug, including dates, quantity and use.

#### 9.5 **Investigational Product Retention at Study Site**

The Investigator (or designee) is responsible for maintaining accurate accountability records of the investigational product throughout the clinical study. All study drug received at the site must be inventoried and accounted for in an accountability log provided by the Sponsor. All dispensing and accountability records will be available for Sponsor review. Study drug accountability will be verified during on-site monitoring visits.

Upon the completion or termination of the study, and upon written authorization from the Sponsor, or its representative, all unused and/or partially used study drug should be returned or destroyed at the investigational site, as specified by Sponsor. It is the Investigator's responsibility to ensure that the Sponsor, or its representative, has provided written authorization that procedures for proper disposal of the study drug have been established, and that appropriate records of the disposal are documented and maintained. No unused study drug may be disposed until fully accounted for by the Sponsor monitor (or designee)

#### 9.6 **Warnings and Precautions**

**Note:** Subjects must not receive any vaccinations from within 2 weeks of screening until Day 56.

#### 9.6.1 **Infusion Reaction**

SYNT001 will be given as an IV infusion over 1 hour. As with all mAbs administered by IV infusion, infusion reactions are possible. In nonclinical testing of SYNT001 in NHPs, clinical observations were limited to infusion reactions due to the immunogenicity of SYNT001 in NHPs. These reactions included transient emesis/vomitus which typically occurred within 1 hour of dosing at all dose groups, but only after the third weekly infusion following the development of ADAs. Transient histamine-type responses were noted 30 minutes post-dose in some animals in all dose groups, but only following the third weekly infusion as above. These reactions were consistent with a histamine reaction (decreased activity, periocular swelling, erythema, facial flushing, eyelids partially/completely closed, and/or generalized weakness). With the exception of vomitus/emesis and red skin discoloration associated with injection or blood draw sites, these observations spontaneously resolved within 1-hour post-dose. Subsequent pretreatment with intramuscular diphenhydramine prevented further histamine-type reactions. All doses of SYNT001 were administered by bolus infusion over approximately 5 minutes in the NHP studies. However, all of the observed infusion reactions (including vomitus/emesis and

histamine-type reactions) associated with ADAs are not at all predictive of what may occur in humans [Bugelski 2004, Ponce 2009] and furthermore, are not considered relevant to predicting responses in humans [ICH S6(R1) 2011].

Typically, infusion reactions to monoclonal antibodies observed in human studies develop within 30 minutes to 2 hours after the initiation of drug infusion, although symptoms may be delayed for up to 24 hours. Most are mild in severity, although severe and even fatal reactions can occur.

# Guidelines for Grading and Management of Allergic or Infusion-Related Reactions

Allergic and/or infusion-related reactions include hypersensitivity reactions and cytokine release syndromes. These reactions are experienced by patients during or within hours of the infusion of monoclonal antibody therapy. Symptoms can include flushing, alterations in heart rate and blood pressure, dyspnea, bronchospasm, back pain, fever, urticaria, edema, nausea, and all types of rashes. Anaphylaxis is recognized as a severe, life-threatening, generalized, or systemic reaction. This is a medical emergency characterized by rapidly developing life-threatening airway and/or breathing and/or circulation problems usually associated with skin or mucosal changes.

Management of Grade 1 infusion reactions include decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen.

Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. See Figure 1 and Figure 2 for details on the management of Grades 1-2 and Grade 3 or higher infusion reactions. The severity of and management of allergic or infusion-related reactions will be graded and managed using NCI CTCAE Version 4.03 (see Table 5).

Figure 1: Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions



If symptoms and signs resolve completely either spontaneously or after administration of diphenhydramine with or without hydrocortisone, consider rechallenge:

Wait at least 20 minutes following medication administration before commencing rechallenge at an infusion rate of 50% or less of the initial infusion rate or

Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction

Syntimmune, Inc.


Amendment 2.0 Final 12 April 2017

Figure 2: Management of Severe (Grade 3 or higher) Infusion Reactions

Subject presents with any of the below:

- Urticaria
- Airway threatened by angioedema
- Angioedema: Lip, mouth, facial swelling
- Respiratory compromise wheezing, dyspnea, stridor or hypoxia (O2 saturation < 90%)
- BP < 90 mmHg SBP or >30% decrease from patient baseline



Start basic life support:

- High oxygen flow
- On bed, head down, legs up
- Large bore IV cannula, 1 L normal saline STAT
- Initiate vital signs at least every 15 minutes



Consider (under medial direction):

Epinephrine 1:1000

• 0.3 mg (0.3 mL) IM into lateral thigh



Airway Threatened: Nebulized epinephrine 1:1000, 3–5 mL (3–5 mg)

**Bronchospasm:** Nebulized salbutamol 5 mg

(Wheeze or Hypoxia) Consider: Intubation / nebulized epinephrine

**Hypotension:** Place on cardiac monitor

(Systolic BP <100 mmHg) Further epinephrine 1:1000, 0.3 mg IM and

IV normal saline bolus 20 mL/kg STAT as needed

Have vasopressin on hand



Transfer to Emergency Room/ICU Observe until all symptoms resolved.

Table 5: Grading and Management of Allergic or Infusion-Related Reactions

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Infusion-<br>Related<br>Reaction | Mild transient<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Allergic<br>Reaction | Transient<br>flushing or<br>rash, drug<br>fever<br>< 38.0°C.<br>Intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Anaphylaxis | - | - | Symptomatic<br>bronchospasm, with or<br>without urticarial;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Cytokine<br>release<br>syndrome | Mild<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>pressor or<br>ventilator<br>support<br>indicated | Death |

Abstracted from NCI CTCAE Version 4.03.

### 9.6.2 Potential Immune Effects

An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels after a single dose and further decreases after multiple doses up to a 70% to 80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within 30% of baseline levels observed at pretreatment occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.

Given the normal adult range of IgG of 500 to 1600 mg/dL (Agarwal and Cunningham-Rundles, 2007; Furst, 2009; Gonzalez-Quintela et al, 2008; Joliff et al, 1982; Keystone et al, 2007; McMillan et al, 1997; van Vollenhoven et al, 2013), with a mean of 1150 mg/dL, a 50% decrease in the mean would be to 575 mg/dL and a 50% decrease from the low end of the normal range used for the inclusion criteria of 600 mg/dL would be to 300 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 120 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency [Ameratunga 2013], the levels will be transient. Further, as reported for other therapies used for pemphigus, the temporary (ie, less than 4 months) depletion of IgG (up to 95% reduction of total IgG as seen with immunoadsorption) does not appear to impart an increased risk of infection (Eming, 2006; Furst, 2009; Keystone et al, 2007; Schmaldienst et al, 2001; van Vollenhoven et al, 2013). Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to reverse the low IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

An antibody blocking FcRn is expected to also down modulate innate and adaptive immunity and the catabolism of IgG-containing immune complexes (IC). Specifically, it is expected that anti-FcRn will promote the clearance of IgG-containing ICs and the effects of these IC on stimulating innate immune cell production of inflammatory cytokines (e.g., IL-12, interferon-γ, and tumor necrosis factor [TNF]) and inhibit the processing and presentation of antigens contained within IC and thus the antigen-specific activation of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells. Therefore, subjects with pre-existing conditions that are dependent upon IgG antibodies, such as chronic infections (e.g., HIV, HBV or HCV), will be excluded from this study, as will subjects with active infection in general.

SYNT001 administration could decrease the level of protective antibodies from prior vaccinations. Protective antibody levels for tetanus and varicella-zoster virus (chickenpox) are to be tested in accordance with Section 6.7.3.

### 10 CONCOMITANT MEDICATION AND TREATMENT

All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted

Use of the following treatments will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine.
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations through Day 56. Following Day 56, subjects may be vaccinated at the discretion of the Investigator.

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

In cases in which concomitant medications are used, details to be recorded include the following: medication name, start date and time, stop date and time, dose, route, frequency, and reason for use. The concomitant medication names are to be coded using the World Health Organization

(WHO) Drug Dictionary (WHO-DD March 2013, Type B2 or later) and classified by anatomical therapeutic chemical (ATC) categories.

### 11 SAFETY

## 11.1 Safety Parameters

Clinical and laboratory AEs will be graded using the NCI CTCAE; Version 4.03 (See Appendix A).

Subjects will be monitored throughout the treatment and follow-up period for occurrence of AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status, vital sign measurements, and laboratory data (including PD). Safety parameters to be measured/assessed include PEs, vital sign measurements, hematology, serum chemistries, urinalysis, and ECG.

### 11.2 Adverse Event Definition

An AE is defined as any untoward medical occurrence in a clinical trial subject associated with the use of a drug, whether considered drug related. An AE can be an unfavorable and unintended sign (e.g., an abnormal laboratory value finding), a symptom, or a disease temporally associated with the use of a drug, without judgment as to causality. An AE can arise from use of the drug (e.g., use in combination with another drug) and from any route of administration, formulation or dose, including an overdose. An AE also includes, but is not limited to, any clinically significant worsening of a pre-existing condition. Examples include:

- Any sign, symptom, physical finding, or laboratory result that has worsened in nature, severity or frequency compared to baseline;
- Reactions from an investigational drug, including those occurring because of an overdose, abuse of the study drug, withdrawal phenomena, sensitivity or toxicity;
- Concurrent illness that was not present or worsens in nature, severity, or frequency compared to baseline;
- Injury or accident; and/or
- Exacerbation of a pre-existing condition.

For data collection, all untoward events that occur after informed consent through the last study visit are to be recorded on eCRFs by the investigational site.

While pregnancy alone is not considered as an AE or SAE, any pregnancy complication(s) should be recorded as an AE(s) or SAE(s) (if applicable). Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions (see below). Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. If a female subject becomes pregnant during the conduct of the study, the Investigator must notify the Sponsor according to the procedures provided in Section 11.3.8).

# 11.3 Evaluating Adverse Events

The Investigator will determine the seriousness, intensity, and causality of an AE associated with the use of the study drug (i.e., events where there is a reasonable possibility that the event may have been caused by the study drug) based on the definitions that follow.

### 11.3.1 Serious Adverse Events

(Notify Medpace Safety within 24 hours; document on eCRF)

The SAE definition and reporting requirements are in accordance with Title 21 Part Code of Federal Regulations (CFR) 312.32 and the Guidance for Industry and Investigators Safety Reporting Requirements for Investigational New Drug (INDs) and Bioavailability /Bioequivalence Studies.

SAE: An AE is considered "serious" if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:

• <u>Death:</u> This includes any death that occurs while the subject is "on study" through the last study visit.

**Note:** Death is an outcome of an AE, and not an AE. The event(s) that caused death (e.g., illness, accident) is the SAE. Death due to any other cause(s) must also be reported as an outcome of the reportable SAE.

- <u>Life-threatening adverse drug event:</u> An AE or suspected adverse reaction is considered "life threatening" if, in the view of either the Investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.
- Inpatient hospitalization or prolongation of existing hospitalization:

In the absence of an AE, the Investigator should not report hospitalization or prolongation of hospitalization. This is the case in the following situations:

- Hospitalization or prolongation of hospitalization is needed for a procedure required by the protocol
- Hospitalization or prolongation of hospitalization is part of routine procedure followed by study center

- Hospitalization for survey visits or annual physicals
- Hospitalization for observation with release within 24 hours

In addition, a hospitalization planned before the start of the study for a pre-existing condition, which has not worsened, does not count as an SAE.

# • Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

- Congenital anomaly/birth defect
- <u>Important medical event:</u> An event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

### 11.3.2 Overdose

An overdose is defined as a significant variation from the recommended/scheduled dosage for a product. The dosing for this study will be conducted in a controlled clinical setting and an overdose is not anticipated. However, in the event of an accident, for this study, an overdose of SYNT001 is considered a dose that is two-fold higher than the intended dose for the subject.

### 11.3.3 Non-Serious Adverse Events

(Document on eCRF)

All other AEs, not fulfilling the previous definitions, are classified as non-serious.

### 11.3.4 Protocol-Related Adverse Events

AEs that are not test drug related may nevertheless be considered by the Investigator or the Medical Monitor to be related to the conduct of the clinical study. That is, the event may be related to the fact that a subject is participating in the study. For example, a protocol-related AE may be an event that occurs during a screening period or that is related to a procedure required by the protocol.

### 11.3.5 Assessment of Causality

A medically qualified Investigator must assess the relationship of any AE (including SAEs) to the use of the investigational product, as related or not related, based on clinical judgment and using all available information, and may include consideration of the following factors:

- Possible alternative causes of the AE, including the disease under treatment, pre-existing conditions, concomitant use of other drugs, and presence of environmental or genetic factors.
- The temporal association between drug exposure and onset of the AE.
- Whether the manifestations of the AE are consistent with known actions or toxicity of the investigational product.
- The AE resolved or improved with decreasing the dose or stopping use of the investigational product (dechallenge). Judgment should be used if multiple products are discontinued at the same time.

The causal relationship between the study medication and the AE will be assessed using one of the following categories:

**Not Related:** Factors consistent with an assessment of Not Related include:

- Temporal relationship is lacking (e.g., the event did not occur within a reasonable time frame following administration of the study medication); or
- Other causative factors more likely explain the event (e.g., a pre-existing condition, other concomitant treatments).

**Related:** Factors consistent with an assessment of Related include:

- There is a positive temporal relationship (e.g., the event occurred within a reasonable time frame following administration of study medication); or
- The AE is more likely explained by the investigational product than by another cause (i.e., the AE shows a pattern consistent with previous knowledge of the investigational product or the class of the investigational product)

#### 11.3.6 **Recording Adverse Events**

All AEs (including SAEs) are to be accurately recorded on the Adverse Event page of the subject's eCRF. The severity of each AE will be graded using the NCI CTCAE, Version 4.03. The date of onset as well as the end date of the event also should be recorded or the event should be entered as "ongoing". In addition, the method used to treat the AE and the outcome of the AE also will be noted. The Investigator will assess the relationship of the event to study drug.

#### 11.3.7 **Planned Hospitalization**

A hospitalization planned by the subject prior to the first dose of study medication is considered a therapeutic intervention and not the result of a new SAE and should be recorded as medical

history. If the planned hospitalization or procedure is executed as planned, the record in the subject's medical history is considered complete. However, if the event/condition worsens during the trial, it must be reported as an AE.

### 11.3.8 Reporting Pregnancies

If a female subject or the female partner of a male subject becomes pregnant during the course of the study, the Investigator must report the pregnancy to the Medpace Safety using the **Pregnancy Reporting Form** within **24 hours** of becoming aware of the event. The Investigator must obtain consent to collect pregnancy information (including the status of the newborn, if applicable).

If some of the information required for completion of the Pregnancy Reporting Form is unavailable at the time of the initial report, follow-up reports will be completed and submitted within 24 hours of becoming aware of the new information. Any pregnancy will be followed through delivery for the observation of any SAEs. Any SAE that occurs during pregnancy must be recorded on the SAE report form in the EDC system (e.g., maternal serious complications, therapeutic or spontaneous abortion, ectopic pregnancy, stillbirth, neonatal death, congenital abnormality, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs (See Section 11.3.9).

### 11.3.9 Serious Adverse Event Reporting

## 11.3.9.1 Governing Regulatory Requirements

Compliance with this request for prompt reporting is essential in that the sponsor is responsible for informing the US Food and Drug Administration (FDA) and other regulatory authorities as well as all other participating Investigators of the event.

Under FDA ruling (US Code of Federal Regulations, Title 21 CFR Part 312.32) and the ICH Guidelines for Clinical Safety Data Management Definitions and Standards for Expedited Reporting, the sponsor is required to submit written documentation, in the form of a safety report, detailing:

- Any event associated with the use of the drug, that is both <u>serious and unexpected</u>, or
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects, including reports of mutagenicity, teratogenicity, or carcinogenicity.

Written submission must be made by the sponsor to the FDA and the IRBs as soon as possible and in no event later than 15 calendar days after the sponsor's initial notification of the event. The sponsor shall also inform all Investigators.

# 11.3.9.2 Time Frame for Reporting

Any death, SAE, pregnancy, or unexpected (and severe) AE experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, , must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee).

Contact information for **SAE** reporting:



Additionally, the Investigator will be able to contact the **Medical Monitor**:



### 11.3.9.3 Information to be Provided by the Investigator

SAEs must be recorded on the SAE form in the EDC system. This requirement includes all SAEs that occur after informed consent through the last study visit.

The minimum information required for SAE reporting includes identity of Investigator, site number, subject number, an event description, SAE term(s), onset date, the reason why the event is serious (i.e., the seriousness criteria) and the Investigator's assessment of the relationship of the event to study treatment. Additional SAE information including medications or other therapeutic measures used to treat the event, action taken with the study treatment due to the event, and the outcome/resolution of the event will be recorded. Paper forms for reporting SAEs will be provided to the study sites as back-up in case the EDC system is not accessible.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. Furthermore, the Investigator may be required to provide supplementary information as requested by Syntimmune or designee.

When reporting an SAE, the following additional points should be noted:

When the diagnosis of an SAE is known or suspected, the Investigator should report the
diagnosis or syndrome as the primary SAE term, rather than as signs or symptoms. Signs
and symptoms may then be described in the event description. For example, dyspnea
should not be used as an SAE term if the diagnosis, which caused the dyspnea, is known
to be malignant pleural effusion.

- Death should not be reported as an SAE, but as an outcome of a specific SAE, unless the event preceding the death is unknown. In the exceptional case where the events leading to death are unknown, then death may be used as an event term. If an autopsy was performed, the autopsy report should be provided.
- While most hospitalizations necessitate reporting of an SAE, some hospitalizations do not require SAE reporting, as follows:
  - Elective or previously scheduled surgery, e.g., a previously scheduled ventral hernia repair
  - Procedures for pre-existing conditions that have not worsened after initiation of treatment
  - Pre-specified study hospitalizations for observation
  - Events that result in hospital stays of less than 24 hours and that do not require admission, e.g., an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics
- SAEs must, however, be reported for any surgical or procedural complication resulting in prolongation of the hospitalization.

### 11.3.10 Regulatory Reporting

Syntimmune (or designee) will process and evaluate all SAEs as soon as the reports are received. For each SAE received, Syntimmune will decide as to whether the criteria for expedited reporting have been met.

Syntimmune (or designee) will submit SAEs that meet the criteria for expedited reporting to the regulatory authorities in accordance with local regulations governing safety reporting. Reporting of SAEs by the Investigator to his or her IRB will be done in accordance with the standard operating procedures and policies of the IRB. Adequate documentation must be maintained showing that the IRB was properly notified.

## 11.3.11 Follow-up Information on a Serious Adverse Event (SAE)

Appropriate diagnostic tests should be performed and therapeutic measures, if indicated, should be instituted. Appropriate consultation and follow-up evaluations should be carried out until the event has returned to baseline or is otherwise explained by the Investigator.

If all required information on the SAE form is not available at the time of the initial report, follow-up information will be completed in the EDC system.

## 11.4 Other Safety Considerations

### 11.4.1 Laboratory Data

All laboratory data obtained during the study should be reviewed. Any abnormal value that leads to a change in subject management (e.g., requirement for additional medication or monitoring) or is of clinical significance by the Investigator should be reported as an AE and/or SAE as appropriate, unless this value is consistent with values obtained before entry into the study.

### 11.4.2 Medication Errors

Any medication error that results in an AE, even if it does not meet the definition of serious, requires reporting within 24 hours to the safety Medical Monitor.

## 11.4.3 Follow-Up of Adverse Events

Any SAE or AE assessed as related to study drug must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. The Investigator will follow all drug related AEs until there is a return to the subject's baseline condition, or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary. The status of all AEs will be documented as of the last study visit.

Where a diagnosis is possible, it is preferable to report this diagnosis rather than a series of terms (signs/symptoms) relating to the diagnosis.

### 11.5 Safety Monitoring for Dose Escalation

Following dosing in each cohort, all safety/tolerability data (e.g., PEs, vital signs [including pulse oximetry], clinical safety laboratory tests, ECGs and AE/SAE assessments) as well as any available and relevant PD data collected through Day 42 will be reviewed by the DEC. A decision to escalate to the next cohort will be made. The recommendation may be to continue to

the next scheduled dose level, discontinue the study or to modify dosing to a dose less than the current dose or higher than the current dose but lower than the next planned dose.

### 12 STATISTICAL CONSIDERATIONS

All descriptive and inferential statistical analyses will be performed using the most recently released and available Statistical Analysis System (SAS) software, unless otherwise noted. Missing data will not be imputed unless otherwise stated. All clinical data captured will be provided in data listings. A Statistical Analysis Plan (SAP) and a Pharmacokinetic Analysis Plan (PAP) will be finalized prior to database lock.

# 12.1 General Design

All data for enrolled subjects will be presented in data listings by subject number.

Continuous data will be described using descriptive statistics: number of observations (n), mean, standard deviation (SD), median, minimum, and maximum. Frequencies and percentages will be used for summarizing discrete (categorical) data. When categorical data are presented, the percent will be suppressed when the count is zero to draw attention to the non-zero counts. The denominator for all percentages, unless otherwise specified, will be the number of subjects in the specified analysis population.

### 12.2 Sample Size Justification

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

### 12.3 Statistical Considerations

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). The SAP may modify the plans outlined in the protocol; any deviations from the previously described statistical plan will be described and justified in an SAP amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate and will be described in the SAP. Methods of handling of missing data for different endpoints will be further specified in the SAP. In general, where individual data points are missing because of insufficient samples, dropouts, or other reasons, the data will be analyzed based on reduced denominators unless specified otherwise in the SAP.

Results will be summarized by cohorts.

## 12.3.1 Study Populations

Three populations will be employed in the analysis of study data:
• The **intent-to-treat (ITT)** population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population.

- The **PK** population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters.
- The **PD** population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the ITT, PK, and PD populations, where appropriate.

## 12.3.2 Subject Accountability, Demographics, and Baseline Characteristics

Subject disposition, demographic information and baseline characteristics will be presented. Any discrepancy between treatment to be given and treatment received will be accounted for in these displays.

#### 12.3.3 Concomitant Medications

Concomitant medications will be coded using WHO Drug Dictionary (WHO-DD March 2013, Type B2 or later) and the data will be summarized and presented in tables and listings.

## 12.4 Planned PK Analysis

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and  $AUC_{0-24}$  and  $AUC_{0-\infty}$ . PK parameters will be determined using noncompartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, SD, coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

For calculation of mean concentrations and generation of mean concentration-time profiles, all below the limit of quantification (BLQ) values will be set to zero except when an individual BLQ falls between 2 quantifiable values, in which case it will be omitted.

If there are values above the BLQ, but too sparse to allow full analysis, descriptive statistics will be performed on available values.

## 12.5 Safety Data

Safety observations and measurements include AEs, safety laboratory tests, vital sign measurements, PEs, and ECGs.

Treatment-emergent AEs will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

AEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject, cohort, and overall per SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by cohort. Incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the local laboratory.

Vital sign measurements and change from baseline will be summarized at each scheduled time point by cohort using descriptive statistics.

Arithmetic mean of parameters from triplicate ECG will be calculated first for each participant at each planned time point. Then summary statistics of ECG test parameters (mean of triplicate) and change from baseline to each post-dose time point will be calculated. Shift tables for ECG test result category change (normal, abnormal, clinically abnormal) from pre-dose to each post-dose time point showing number and percentage of subjects with movement between categories will be presented by treatment group. Frequency and percentage of subjects experiencing potential QTc prolongation (QTcF > 450) will be summarized at each time point by cohort.

#### 12.6 Pharmacodynamic/Activity Data

PD results will be summarized by cohort.

## 12.7 Immunogenicity Data

Immunogenicity results will be summarized by cohort.

## 12.8 Interim Analysis

No interim analysis is planned. Safety results will be examined for making dose-escalation decisions; no statistical analyses are planned for aiding these dose-escalation decisions.

## 13 DATA QUALITY ASSURANCE

All data will be entered in a validated electronic data capture system using single data entry. Standard procedures (including following data review guidelines, manual clinical review based on subject profiles, computerized validation to produce queries, and maintenance of an audit file which includes all database modifications) will be followed to ensure accurate data. Clinical personnel will review all data listings for outliers, data inconsistencies, and spelling errors.

During the study, a study site monitor will make site visits to review protocol compliance, compare electronic case report forms (eCRFs) against individual subject medical records, assess drug accountability, and ensure that the study is being conducted using pertinent regulatory requirements. eCRF entries will be verified with source documentation. The review of medical records will be performed in a manner to ensure that subject confidentiality is maintained. Checking the eCRFs for completeness, clarity and cross checking with source documents is required to monitor the progress of the study. Direct access to source data is also required for inspections and audits, and will be carried out giving due consideration to data protection and medical confidentiality. Each Investigator will have assured Syntimmune of full access to complete source data for study participants and associated necessary support at all times.

In addition to routine monitoring procedures, audits of clinical research activities in accordance with standard operating procedures (SOPs) may be performed to evaluate compliance with the principles of GCP. A regulatory authority may also wish to conduct an inspection (during the study or even after its completion). If a regulatory authority requests an inspection, the Investigator must immediately inform Syntimmune that this request has been made. Study conduct may be assessed during the study by a Clinical Quality Assurance representative(s) to ensure that the study is conducted in compliance with the protocol. This designee, as well as the site monitor, will be permitted to inspect the study documents (study protocol, eCRFs, investigational product accountability, original study-relevant medical records). All subject data will be treated confidentially. During the clinical study, access will be available to Syntimmune or their designee (e.g., contract research organization [CRO]) to view the eCRFs after completion of the individual sections of the study. Furthermore, the study protocol, each step of the data-recording procedure and the handling of the data as well as the study report may be subject to independent review by a Quality Assurance representative. Clinical site and study audits will be conducted as necessary to assure the validity of the study data.

#### 14 STUDY ADMINISTRATION

## 14.1 Study Administrative Structure

The study administration structure is provided in Table 6.

**Table 6:** Study Administrative Structure



## 14.2 Ethical Conduct of the Study

The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH E6 Tripartite Guideline (January 1997), and in general, be conducted in a manner consistent with the principles described in the Declaration of Helsinki. The Investigator will ensure that the conduct of the study complies with the basic principles of GCP as outlined in the current version of 21 CFR, subpart D, Part 312, "Responsibilities of Sponsors and Investigators", Part 50, "Protection of Human Subjects", and Part 56, "Institutional Review Boards".

## 14.3 Informed Consent (ICF)

A properly executed, written informed consent document, in compliance with 21 CFR, Part 50 and the ICH guidelines, will be obtained from each subject before the subject is entered into the study and before any study screening procedure is performed that involves risk. Attention will

Pemphigus

be directed to the basic elements required for incorporation into the informed consent under US Federal Regulations for Protection of Human Subjects (21 CFR 50.25[a]) and (21 CFR 50.25[b]), as necessary.

Sample ICFs will be supplied to each site. Syntimmune or its designee must review any proposed deviations from the sample ICF. The final IRB-approved document must be provided to Syntimmune for regulatory purposes.

It is the responsibility of the Investigator, or a person designated by the Investigator, to obtain written informed consent from each subject (or the subject's legally authorized representative) participating in this study after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study. In the case where the subject is unable to read, an impartial witness should be present during the entire informed consent discussion. After the subject has orally consented to participation in the trial, the witness' signature on the form will attest that the information in the consent form was accurately explained and understood. A copy of the ICF must be provided to the subject or to the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

The eCRF for this study contains a section for documenting informed subject consent, and this must be completed appropriately. Signed ICFs must remain in each subject's study file and must be available for verification by site monitors at any time. If new safety information results in significant changes in the risk/benefit assessment, the consent form should be reviewed and updated as necessary. All subjects (including those already being treated) should be informed of the new information, should be given a copy of the revised form, and should give their consent to continue in the study.

#### 14.4 Institutional Review Board

This study is being conducted under US IND 128152. This protocol (and any modifications) and appropriate consent procedures must be reviewed and approved by an IRB. This board must operate in accordance with the current federal or local regulations. The Investigator will send a letter or certificate of IRB approval to Syntimmune (or designee) before subject enrollment and whenever subsequent modifications to the protocol are made.

## 14.5 Dose Escalation Committee

The DEC will be responsible for confirming the safety of the investigative product prior to dose escalation, as well as the dose level for each successive cohort. In addition, over the course

of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects. The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions.

## 14.6 Future Use of Subject Samples

Not all the tissue and blood components obtained during this study may be required for the tests that are part of the clinical trial. Available samples may be used for additional research. This research will help to understand disease subtypes, drug response and AE, and possibly identify new drug targets or biomarkers that predict subject response to treatment. The use of the samples for internal research will be done using the guidelines defined by the FDA guidance for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individual Identifiable (issued 25 April 2006) and the European Medicines Agency (EMA) Reflection Paper on Pharmacogenetic Samples, Testing and Data Handling (Doc. Ref.

EMEA/CHMP/PGxWP/201914/2006; 15 November 2007). If a subject requests destruction of their tissue and blood samples and the samples have not yet been de-identified, Syntimmune will destroy the samples as described in this FDA guidance. Syntimmune will notify the Investigator in writing that the samples have been destroyed.

#### 15 CONDITIONS FOR MODIFYING THE PROTOCOL

Protocol modifications to ongoing studies must be made only after consultation between a Syntimmune representative and the Investigator. Protocol modifications will be prepared, reviewed, and approved by Syntimmune representatives.

All protocol modifications must be submitted to the IRB for information and approval in accordance with local requirements, and to regulatory agencies if required. Approval must be obtained before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to study subjects, or when the change involves only logistical or administrative aspects of the trial (e.g., change in site monitor, change of telephone number).

## 16 CONDITIONS FOR TERMINATING THE STUDY

Syntimmune has the right to terminate the study at any time. In terminating the study, Syntimmune and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests.

## 17 STUDY DOCUMENTATION, CRFS, AND RECORD KEEPING

## 17.1 Investigator's Files and Retention of Documents

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into 2 separate categories as follows: (1) Investigator's study file and (2) subject clinical source documents.

The Investigator's study file will contain the protocol and protocol amendments, eCRFs, query forms, IRB and governmental approval with correspondence, sample informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

Subject clinical source documents (usually predefined by the project to record key efficacy and safety parameters independent of the eCRFs) may include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, electroencephalogram, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject screening and enrollment logs. The Investigator must keep these 2 categories of documents on file for at least 2 years following the marketing application approval date for the study treatment and for the indication being investigated or for 2 years after the development program is discontinued and the FDA notified. After that period, the documents may be destroyed subject to local regulations with prior written permission from Syntimmune. If the Investigator wants to assign the study records to another party or move them to another location, Syntimmune must be notified in advance.

If the Investigator cannot guarantee the archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and Syntimmune to store these in a sealed container outside of the study site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storing outside of the study site.

## 17.2 Source Documents and Background Data

Investigators must maintain adequate and accurate source documents on which the eCRFs for each subject are based. They are separate and distinct from the eCRFs.

These records include detailed notes on the following:

- Medical history
- Date and time of informed consent with Health Insurance Portability and Accountability
  Act (HIPAA) authorization either contained in the ICF or presented to the subject
  candidate as a standalone document
- Description of the complete consenting process
- The basic identifying information that linked the subject's medical record with the eCRFs
- The results of all diagnostic tests performed, diagnoses made, therapy provided, and any other data on the condition of the subject
- The medical condition of the subject during their involvement in the study
- All AEs
- The subject's exposure to the study medication
- The subject's exposure to any concomitant therapy
- All relevant observations and data on the condition of the subject throughout the trial
- Justification for all entries in the subject's eCRF

A subject log of all potentially eligible subjects considered, but not consented, for obvious deviations from the entry criteria, will be kept at each site. The log will contain subjects' initials, diagnosis, eligibility, or, if not eligible, reason for not consenting. All consented subjects will be logged, regardless of whether they ultimately enroll.

Upon request, the Investigator will supply Syntimmune with any required background data from the study documentation or clinic records. This is particularly important when eCRFs are illegible or when errors in data transcription are suspected. In case of special problems or governmental queries or requests for audit inspections, it is also necessary to have access to the complete study records, provided that subject confidentiality is protected.

#### 17.3 Audits and Inspections

The Investigator should understand that source documents for this study should be made available to appropriately qualified personnel from Syntimmune (or designee), or to health authority inspectors after appropriate notification. The verification of the eCRF data must be by direct inspection of source documents.

## 17.4 Electronic Case Report Forms

Clinical trial data for this study will be captured on eCRF designed for computer processing and analysis. This computerized system will be validated and compliant with 21 CFR Part 11. Corrections to data will be made using 21 CFR Part 11, Electronic Records; Electronic Signatures. If corrections are made after review and sign-off by the Investigator, he/she must be aware of the changes and provide written acknowledgement. There will also be an electronic audit trail. Corrections on paper CRFs must be initialed and dated by the person making the change. The Investigator agrees to provide all information requested on the eCRF in an accurate manner using instructions provided. The Investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported to Syntimmune in the eCRF and in all required reports.

An eCRF is required to be submitted for every subject who receives any amount of study drug. This includes submission of retrievable data on subjects who withdraw before completion of the study. Prior to submission, eCRFs must be reviewed for completeness and accuracy, and signed and dated where either indicated, by the Principal Investigator or authorized delegate from the study staff. If a subject stops treatment or terminates from the study, the dates and reasons must be noted on the eCRF.

# 18 MONITORING THE STUDY

It is understood that the responsible Syntimmune site monitor (or designee) will contact and visit the Investigator regularly and will be allowed on request to inspect the various records of the trial (eCRFs and other pertinent data) if subject confidentiality is maintained in accordance with local requirements.

It will be the site monitor's responsibility to inspect the eCRFs at regular intervals throughout the study, to verify the adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The site monitor should have access to laboratory test reports and other subject records needed to verify the entries on the eCRF. The Investigator (or designee) must agree to cooperate with the site monitor to ensure that any problems detected during these monitoring visits are resolved.

#### 19 CONFIDENTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECORDS

The Investigator must ensure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On eCRFs or other documents submitted to Syntimmune, subjects should be identified by an identification code and not by their names. The Investigator should keep a subject enrollment log showing codes, names, and addresses. The Investigator should maintain documents not for submission to Syntimmune (e.g., subjects' written consent forms) in strict confidence.

Authorized regulatory officials and Syntimmune personnel (or their representatives) will be allowed full access to inspect and copy the records. All study drugs, subject bodily fluids and tissue, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by Syntimmune.

The Principal Investigator also agrees that all information received from Syntimmune, including but not limited to the IB, this protocol, eCRFs, the INDs, and any other study information remain the sole and exclusive property of Syntimmune during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from the sponsor. The Principal Investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 20 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. The Investigator agrees that any manuscript or abstract they author may be published only after receiving written permission from Syntimmune.

If Syntimmune coordinates a publication or presentation of study results from all study sites, the participation of Investigator or other representatives of study site as a named author shall be determined in accordance with Syntimmune policy and generally accepted standards for authorship.

#### 21 REFERENCES

Agarwal S and Cunningham-Rundles C. Assessment and clinical interpretation of reduced IgG values. Ann Allergy Asthma Immunol. 2007;99:281-283.

Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID), which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. *Clin. Exp. Immunol.* 2013;174: 203-211.

Bugelski PJ and Treacy G. (2004) Predictive power of preclinical studies in animals for the immunogenicity of recombinant therapeutic proteins in humans. *Curr Opin Mol Ther*. 2004;6:10–16.

Eming R, Hertl M. Immunoadsorption in pemphigus. Autoimmunity. 2006;39:609-616.

Furst DE. Serum immunoglobulins and risk of infection: how low can you go? Semin Arthritis Rheum. 2009;39:18-29.

Gonzalez-Quintela A, Alende R, Gude R, Campos J, Rey J, Meijide LM, Fernandez-Merino C, Vidal C. Serum levels of immunoglobulins (IgG, IgA, IgM) in a general adult population and their relationship with alcohol consumption, smoking, and common metabolic abnormalities. Clin Exp Immunol. 2008;151:42-50.

International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) (2011). S6(R1) Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals. Accessed 03 June 2016.

http://www.ich.org/products/guidelines/safety/safety-single/article/preclinical-safety-evaluation-of-biotechnology-derived-pharmaceuticals.html

Joliff CR, Cost KM, Stivrins PC, Grossman PP, Nolte CR, Franco SM, et al. Reference intervals for serum IgG, IgA, IgM, C3 and C4 as determined by rate nephelometry. Clin Chem. 1982;28:126-128.

Keystone E, Fleischmann R, Emery P, Furst DE, van Vollenhoven R, Bathon J, et al. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007;56:3896-3908.

McMillan SA, Douglas JP, Archbold GPR, McCrum EE, Evans AE. Effect of low to moderate levels of smoking and alcohol consumption on serum immunoglobulin concentrations. J Clin Pathol. 1997;50:819-822.

Nixon AE, Chen J, Sexton DJ, Muruganandam A, Bitonti AJ, Dumont J, Viswanathan M, Martik D, Wassaf D, Mezo A, Wood CR, Biedenkapp JC, TenHoor C. (2015). Fully human monoclonal antibody inhibitors of the neonatal Fc receptor reduce circulating IgG in non-human primates. Front. Immun. 6:176

Ponce R, Abad L, Amaravadi, L, et al. Immunogenicity of biologically-derived therapeutics: assessment and interpretation of nonclinical safety studies. *Regul Toxicol Pharmacol*. 2009;54,164–182.

Roopenian, D.C., Christianson, G.J., Sproule, T.J., Brown, A.C., Akilesh, S., Jung, N., Petkova, S., Avanessian, L., Choi, E.Y., Shaffer, D.J., Eden, P.A., Anderson, C. L. The MHC class I-like IgG receptor controls perinatal IgG transport, IgG homeostasis, and fate of IgG-Fc-coupled drugs. 2003. J. Immun. 170 3528-3533

Schmaldienst S, Müllner M, Goldammer A, Spitzauer S, Banyai S, Hörl WH, Derfler K. Intravenous immunoglobulin application following immunoadsorption: benefit or risk in patients with autoimmune disease? Rheumatology. 2001;40:513-521.

van Vollenhoven RF, Emery P, Bingham CO 3rd, Keystone EC, Fleischmann RM, Furst DE, et al. Long-term safety of rituximab in rheumatoid arthritis: 9.5-year follow-up of the global clinical trial programme with a focus on adverse events of interest in RA patients. Ann Rheum Dis. 2013;72:1496-502.

Appendix A: NCI CTCAE, Version 4.03

# Appendix B: Pemphigus Disease Area Index (PDAI)

## Pemphigus Disease Area Index (PDAI)

| Skin | Activity | | Damage |
|---|---|---|---|
| Anatomical Locatio | • | | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion |
| | 0 absent 1 1-3 lesions, up to one >2 cm in any diameter, none > 6 cm 2 2-3 lesions, at least two > 2 cm diameter, none > 6 cm 3 >3 lesions, none > 6 cm diameter 5 >3 lesions, and/or at least one >6 cm 10 >3 lesions, and/or at least one lesion >16 cm diameter or entire area | | 0 absent<br>1 present |
| Ears | | | |
| Nose | | | |
| Rest of the face | | | |
| Neck | | | |
| Chest | | | |
| Abdomen | | | |
| Back, buttocks | | | |
| Arms | | | |
| Hands | | - | |
| Legs | | - | |
| Feet | | | |
| Genitals | 400 | | /12 |
| Total skin | /120 | | 112 |
| Scalp | <b>-</b> | | Doct inflammaton |
| Scalp | Erosion/Blisters or new erythema | | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion |
| | 0 absent 1 in one quadrant 2 two quadrants 3 three quadrants 4 affects whole skull 10 at least one lesion > 6 cm | | 0 absent<br>1 present |
| Total Scalp (0-10) | /10 | | /1 |
| Mucous mer | nbrane | | |
| Anatomical<br>Location | Erosion/Blisters | | |
| | 0 absent<br>1 1 lesion<br>2 2–3 lesions<br>5 >3 lesions or 2 lesions >2 cm<br>10 entire area | Number<br>lesions<br>if ≤ 3 | |
| Eyes | | | |
| Nose | | | |
| Buccal mucosa | | | |
| Hard palate | | $\vdash$ | |
| Soft palate | | $\vdash$ | |
| Upper gingiva | | $\vdash$ | |
| Lower gingiva | | $\vdash$ | |
| Tongue | | $\vdash$ | |
| Floor of mouth | | + | |
| Labial bucosa | | $\vdash$ | |
| Doctorior phoney | | | |
| Posterior pharynx | | | |
| Anogenital Total Mucosa | /120 | | |

Copyright ©2007 University of Pennsylvania; All Rights Reserved.

# Syntimmune, Inc.

## SUMMARY OF CHANGES TO CLINICAL STUDY PROTOCOL

# A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

**Medical Monitor:** PPD

43 Thorndike Street, Cambridge, MA 01240

Phone: PPD extension PPD

Mobile: PPD

**Date of Protocol:** Original, 18 January 2017

 Amendment 1.1
 21 March 2017

 Amendment 2.0
 12 April 2017

## **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

#### **SUMMARY**

The SYNT001-103 protocol has been amended under version 2.0 as follows:

- Lengthened subject follow-up to include study visits at Day 84 and Day 112 to follow pharmacodynamics (Serum IgG) and clinical effects out to 12 weeks from the last dose of SYNT001
- Added immune phenotyping to Day 56 assessments
- Contraception requirement in Inclusion and Exclusion criteria updated to correspond to additional study visits (out to Study Day 112; 12 weeks following last dose of SYNT001) for both females and males
- Total blood draw for subjects completing the study at Day 112 updated to approximately 381 mL from 311 mL in Section 6.7
- Allowing vaccinations at the discretion of the Investigator after Day 56
- AE reporting timelines updated to correspond to additional study visits
- Clarifying language for Tetanus and Varicella-Zoster Virus antibody testing follow-up,
   specifying the actual study visit Days when additional testing will be performed
- Clarifying language for Investigator removal of subjects from study to not require consultation with Medical Monitor but to allow it if desired
- Clarifying language for dose escalation stopping rules; rules for stopping escalation are not changed
- Additional text related to potential immune effects and corresponding references added
- Various typographical and formatting corrections as well as corrections for consistency made throughout the document.

#### **SPECIFIC CHANGES**

Text deletions are shown using strike through font; new text added in *italic font*.

#### **SECTION 1, STUDY SYNOPSIS**

In addition to the changes in the section below, the synopsis has been updated to reflect all changes in the body of the protocol.

#### Duration of subject participation and duration of study

• Up to 70-126 days (40 18 weeks): Screening of up to 2 weeks (14 days); Treatment dosing period of 8 weeks (56 days) 28 days; Follow-up period of and 4 8 weeks (56 28 days)

#### Table 1, Schedule of Assessments

- Table updated to show Treatment Period spanning Day 0 through Day 56
- Table updated to show Follow-up Period spanning Day 84 through Day 112
- Table updated by adding a Day 84 visit and a Day 112/ Early Termination visit, with associated assessments described in Section 7
- Adverse Events and Concomitant Medications:
  - To be collected from the date that the ICF was signed through the last study visit until 28 days after the last dose of study drug

#### • Footnote d: Clinical safety labs:

O Hematology, clinical chemistry, and urinalysis (see Section 6.6 for a complete list). Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 11256. PD biomarkers (albumin levels, hematocrit, hemoglobin, platelet count, reticulocyte count, LDH, and total and direct bilirubin) will be derived from the clinical safety laboratory results.

## Footnote e: Pregnancy Test:

To be performed at time of screening, prior to first dose of SYNT001 on Day 0
 and on Days 56 and 112 (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing.)

Syntimmune, Inc.  12 April 2017

## • Footnote g: Serology:

Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at *Day 841* month after the Follow Up visit (approximately 2 months after the subject's last dose); if still below the baseline value (or level of detection), the subject will be re-tested at *Day 112* after another month (3 months after last dose). Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level *by Day 112* on Day 56 and upon 2 retests (2 and 3 months following last dose of SYNT001), will be referred to their primary care physician for further management. See Section 6.7.3 for additional information.

## • Footnote i: Immunogenicity:

- Blood samples will be collected pre-dose when collected on dosing days.
   Samples will be collected on Days 0, 14, 28, 56, 84 and 112. See Section 6.7.6 for additional information.
- Footnote q: Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management. Extended follow-up visits will occur only if additional testing for anti-tetanus and/or anti-VZV titers are required. These visits will occur as needed at approximately 2 months post last dose and 3 months post last dose.

#### **SECTION 4 STUDY DESIGN**

### Section 4.3, Overview of Study Design

- On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, and 56, 84, and 112. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.
- Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42 and 5642 for safety assessments, study drug dosing, sample collections, and other study procedures.
- Subjects also will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management. 56 (28 days after receiving their last dose of study drug) for an End of Study/Follow Up visit.
- **Note**: No vaccinations may be given from within 2 weeks of screening *through Day 56*. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator. until 2 months following the last dose of study drug

#### **SECTION 5 STUDY POPULATION**

#### **Section 5.1, Target Population**

• This study will be conducted in approximately 16 male and female subjects (2 cohorts of 8 subjects each) with a confirmed diagnosis of pemphigus (vulgaris or foliaceus); however, a third cohort of up to 8 subjects may be added. Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled visits28 days after last dose. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects may be enrolled with pemphigus foliaceus.

## Section 5.2, Inclusion Criteria

7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from

Syntimmune, Inc.  12 April 2017

- the Screening Period through 30 days after the final dose of study visit drug: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final dose of study visit drug.

#### **SECTION 6 STUDY PROCEDURES**

### Section 6.6, 12-Lead Electrocardiogram (ECG)

• Digital 12-lead ECG measurements will be obtained at screening, on Days 0 and 28 at 5 minutes after the completion of the infusion and at the Day 56 (Follow up) visit. Subjects who conduct their Day 12 visit at the investigative site, as opposed to an athome nurse visit, will have an additional ECG performed. ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each 1–2 minutes apart. See Table 2 for timing window allowances with respect to performing ECG.

#### **Section 6.7, Clinical Laboratory Measurements**

- Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and anti-drug antibody samples) will be performed using established methods by a central laboratory. Safety laboratory panels are defined as listed in Table 3. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and anti-drug antibody samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 11256. The total blood draw for each subject who completes the study at Day 11256, will be approximately 311 381 mL. Please refer to the Laboratory Manual for more information.
- Table 3: Clinical Laboratory Panels, Hematology
  - o CBC with differential and blood smear

## **Section 6.7.1 Pregnancy Testing**

• Pregnancy testing will be performed for women of childbearing potential at screening and prior to first dose of SYNT001 on Day 0 and Days 56 and 112 (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing.)

## Section 6.7.3. Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

• Samples for serum tetanus antibody and Varicella-Zoster virus antibody testing are to be collected at baseline (pre-dose, Day 0) and on Day 56 (Follow-Up visit). Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. Specifically, if the baseline VZV titer is above the detectable level, but Tetanus is not, only the VZV antibody titer will be tested on Day 56. If the Day 56 results are below the baseline value, defined as greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 841 month after the Follow Up visit (approximately 2 months after the subject's last dose); if still below the baseline value (or level of detection), the subject will be re-tested at Day 112after another month (3 months after last dose). Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112on Days 56 and upon 2 retests (2 and 3 months following last dose of SYNT001), will be referred to their primary care physician for further management

# Section 6.7.5 Pharmacodynamic (PD) Sampling

Table 1: Pharmacodynamic/ Activity Assessments

| Parameter | Collection Timepoints |
|---|---|
| IgG, IgG subtypes (IgG1-4), IgA, IgM | Screening, and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, 56, 84 and 11256. |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84 and 11256 |
| • Albumin | Screening, and Days 0, 7, 14,21, 28, 33, 42, 56, 84 and 11256 |
| Anti-Dsg (1 and 3) antibody titer | Screening, Days 0, 7, 14, 33, 56, 84 and 112 <del>56</del> |
| <ul> <li>Complement component 3 (C3)</li> <li>Anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence</li> </ul> | Days 0, 14, 33, 56, 84 and 112 <del>56</del> |
| Exploratory biomarker (RNAseq, Urine IgG) | Days 0, 14, 33, 56, 84 and 112 <del>56</del> |
| Immune phenotyping by flow cytometry for<br>measurement of CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T,<br>monocytes, NK cells and B cells | Days 0, 28 and 2856 |
| Exploratory biomarker (FCGR2A SNP) | Day 0 |

Alexion Confidential

#### **Section 6.7.6 Immunogenicity Testing**

• Up to 4 sSerum samples will be collected for immunogenicity analyses. Samples will be collected on Days 0 (pre-dose), 14, 28, 56, 84 and 56112

#### **Section 6.9 Prior and Concomitant Medication**

 All medications a subject receives within 14 days prior to enrollment through the end of the study (Day 56) will be documented on the source document and eCRF.

Note: No vaccinations may be given from within 2 weeks of screening *through Day 56*. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator. until 2 months following the last dose of study drug.

#### **Section 6.10 Adverse Events Assessments**

• Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form *and is continuing through the last study visit* throughout their participation in the study, including a period of 28 days after study drug dosing. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE

## Section 6.11 Photographs

• On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84 and 11256. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

## **Section 6.12 Skin Biopsies**

• Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33, *56* and *8456* to analyze SYNT001 levels

#### **SECTION 7 STUDY ASSESSMENTS**

#### Section 7.7 Dose 2 Follow-up Day 12

• On Day 12 ( $\pm$  6 hours) the subject *may* will return to the clinic, or be visited by an athome nurse, and the following procedures are to be performed:

## Section 7.11 Treatment Day 28 (Dose 5)

• On Day 28 (± 6 hours 1 Day), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

## Section 7.15 Follow-up Day 42

• PDAI Score (Section 6.4)

## Section 7.16 Follow-up Day 56 (End-of-Study) or Early Termination Visit

- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the sitting position) (Section 6.66.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - *Immune phenotyping*

## Section 7.17 Follow-up Day 84

On Day 84 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Serum tetanus antibody and VZV antibody testing if required. See Section 6.7.3 for additional information.
- *Immunogenicity sample collection (Section 6.7)*

Syntimmune, Inc.  12 April 2017

- PDAI Score (Section 6.4)
- *PD sample collection (Section 6.7)* 
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## Section 7.18 Follow-up Day 112 (End-of-Study) or Early Termination Visit

On Day 112 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody testing if required. See Section 6.7.3 for additional information.
- *Immunogenicity sample collection (Section 6.7)*
- PDAI Score (Section 6.4)
- *PD sample collection (Section 6.7)* 
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)

• AE assessment (Section 6.10)

## **Section 7.16 Extended Follow-up Visits**

• Extended follow-up visits will occur only if additional testing for anti-tetanus and/or anti-VZV titers are required. These visits will occur as needed at approximately 2 months post last dose and 3 months post last dose. See Section 6.7.3.

#### SECTION 8 REMOVING SUBJECTS FROM STUDY

#### **Section 8.3 Replacements**

Subjects withdrawn for a reason other than an AE will be replaced if they have not been
dosed or have only received 1 dose of study drug at the time of discontinuation, up to one
subject per cohort. Subjects who do not receive all doses of study drug will continue to be
followed through all scheduled study visits28 days after their last dose.

## **Section 8.4.1 Dose-Escalation Stopping Rule**

• Dose escalation decisions will be made by a Dose Escalation Committee (DEC) and will be based on safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities, AEs, SAEs, and total IgG levels.

Dose-limiting toxicity (DLT) will be defined generally as elinically significant, severe (Grade 3) AEs occurring in  $\geq 2$  subjects that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and no further dose-escalation to a higher dose will not occur. If the dose-escalation stopping rule is met in during cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics will be reviewed and the cohort may resume (if applicable) or a new a cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met in after Cohort 1, dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met in for the first time during Cohort 2, all safety data and all available pharmacodynamics will be reviewed and the cohort may resume (if applicable) or a new a cohort may be added at a dose a minimum of 30% lower than the Cohort 2 dose. If the stopping rule is not met in after Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data.

## Section 8.4.3 Individual Stopping Rule

• Dosing for any individual subject will be discontinued (i.e., no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator and (following consultation with the Medical Monitor, if desired) suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject may will be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus

#### **SECTION 9 STUDY DRUG**

#### **Section 9.6 Warnings and Precautions**

• **Note:** Subjects must not receive any vaccinations from within 2 weeks of screening until 2 months after the last dose of study drug Day 56.

#### **Section 9.6.2 Potential Immune Effects**

- An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels after a single dose and further decreases after multiple doses up to a 70%-80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within 30% of baseline levels observed at pretreatment normal limits-occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.
- Given the normal adult range of total IgG of 700500-1600 mg/dL (Agarwal and Cunningham-Rundles, 2007; Furst, 2009; Gonzalez-Quintela et al, 2008; Joliff et al, 1982; Keystone et al, 2007; McMillan et al, 1997; van Vollenhoven et al, 2013in some references), with a mean of 1150 mg/dL, a 50% decrease in the mean would be to 575 mg/dL and a 50% decrease from the low end of the normal range used for the inclusion criteria of 700600 mg/dL in this study would be to 350300 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 140120 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency [Ameratunga 2013], the levels will be transient. Further, in other conditions, the temporary (ie, less than 4 months) depletion of IgG (up to 95% reduction of total IgG as seen with immunoadsorption) does not appear to impart an increased risk of infection (Eming, 2006; Furst, 2009; Keystone et al, 2007; Schmaldienst et al, 2001; van Vollenhoven et al, 2013). Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to reverse the low IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

#### SECTION 10 CONCOMITANT MEDICATION AND TREATMENT

- Any medications a subject receives within 14 days prior to enrollment through the end of study (Day 56) will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications maywill result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted.
- Use of the following treatments will not be permitted during the study unless otherwise specified:
  - Rituximab or other anti-CD20 antibody
  - Monoclonal antibodies other than study drug
  - Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine.
  - Topical steroids
  - Any dietary herbal supplements
  - Any investigational drug or device
  - Any vaccinations through Day 56. Following Day 56, subjects may be vaccinated at the discretion of the Investigator.

#### **SECTION 11 SAFETY**

#### **Section 11.2 Adverse Event Definition**

 For data collection, all untoward events that occur after informed consent through the last study visit 28 days after study drug dosing are to be recorded on eCRFs by the investigational site

#### **Section 11.3.1 Serious Adverse Events**

• <u>Death:</u> This includes any death that occurs while the subject is "on study" through the last study visit as well as any death that occurs within 28 days after study drug administration

#### Section 11.3.9.2 Time Frame for Reporting

Any death, SAE, pregnancy, or unexpected (and severe) AE experienced by the subject
after informed consent through the last study visit or within 28 days of receiving study
drug, regardless of relationship to study drug, or any death that occurs more than 28 days
after receiving study drug, and is believed to be study drug related, must be promptly
reported (within 24 hours of the Investigator becoming aware of the event) by telephone
or electronic transmission to the sponsor (or designee)

#### Section 11.3.9.3 Information to be Provided by the Investigator

SAEs must be recorded on the SAE form in the EDC system. This requirement includes
all SAEs that occur after informed consent through the last study visit and through
28 days after study drug dosing, and in addition, any SAE that are assessed as related to
study treatment by the Investigator, even if the SAE occurs more than 28 days after study
drug dosing.

## **Section 11.4.3 Follow-up of Adverse Events**

• Any SAE or AE assessed as related to study drug that led to treatment discontinuation (including clinically significant abnormal laboratory values that meet these criteria) and ongoing 28 days after study drug dosing must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. This follow up guidance also applies to related SAE that occur more than 28 days after study drug dosing. The status of all other continuing AEs will be documented as of 28 days after study drug dosing. The Investigator will follow all subjects who experience drug related AEs until there is a return to the subject's baseline condition, or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary. The status of all AEs will be documented as of the last study visit.

#### **REFERENCES** – The following were added:

Agarwal S and Cunningham-Rundles C. Assessment and clinical interpretation of reduced IgG values. Ann Allergy Asthma Immunol. 2007;99:281-283.

Eming R, Hertl M. Immunoadsorption in pemphigus. Autoimmunity. 2006;39:609-616.

Furst DE. Serum immunoglobulins and risk of infection: how low can you go? Semin Arthritis Rheum. 2009;39:18-29.

Gonzalez-Quintela A, Alende R, Gude R, Campos J, Rey J, Meijide LM, Fernandez-Merino C, Vidal C. Serum levels of immunoglobulins (IgG, IgA, IgM) in a general adult population and their relationship with alcohol consumption, smoking, and common metabolic abnormalities. Clin Exp Immunol. 2008:151:42-50.

Syntimmune, Inc.  12 April 2017
Joliff CR, Cost KM, Stivrins PC, Grossman PP, Nolte CR, Franco SM, et al. Reference intervals for serum IgG, IgA, IgM, C3 and C4 as determined by rate nephelometry. Clin Chem. 1982;28:126-128.

Keystone E, Fleischmann R, Emery P, Furst DE, van Vollenhoven R, Bathon J, et al. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007;56:3896-3908.

McMillan SA, Douglas JP, Archbold GPR, McCrum EE, Evans AE. Effect of low to moderate levels of smoking and alcohol consumption on serum immunoglobulin concentrations. J Clin Pathol. 1997;50:819-822.

Schmaldienst S, Müllner M, Goldammer A, Spitzauer S, Banyai S, Hörl WH, Derfler K. Intravenous immunoglobulin application following immunoadsorption: benefit or risk in patients with autoimmune disease? Rheumatology. 2001;40:513-521.

van Vollenhoven RF, Emery P, Bingham CO 3rd, Keystone EC, Fleischmann RM, Furst DE, et al. Long-term safety of rituximab in rheumatoid arthritis: 9.5-year follow-up of the global clinical trial programme with a focus on adverse events of interest in RA patients. Ann Rheum Dis. 2013;72:1496-502.

# **SYNTIMMUNE**

10-May-2017

**Protocol Number:** 

SYNT001-103

**IND Number:** 

132727

Study Drug:

SYNT001

Protocol Version, Date:

2.0, 12-April-2017

Clarification Letter Version:

1.0

Subject:

**Buccal swab for DNA testing** 

## To Whom It May Concern:

The purpose of this letter is to clarify any question as to the method used for the collection of a subject sample to evaluate a FcGR2A SNP (single nucleotide polymorphism) from clinical protocol SYNT001-103, titled "A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)." The protocol includes an exploratory objective to evaluate FcGR2a SNP as an exploratory biomarker. This objective will be evaluated through the collection of a single buccal swab, from which DNA will be extracted and analyzed. This buccal swab will be collected from the subject prior to dosing on the day of first dose of SYNT001.

The protocol does not specify the collection will be made via buccal swab; however, the laboratory manual provides detailed instructions to the site on the collection materials and methods to be used. Subjects are informed of the assessment and the means by which it will be collected and data generated from it in the Informed Consent Form. In the event that there is a future protocol amendment, this clarification will be incorporated.

| Sincerely. | טאי |
|------------|-----|
| Syntimmune | Inc |

257 Park Ave S, 15th Floor, New York, New York, 10010

## SYNTIMMUNE

11-Aug-2017

Protocol Number: SYNT001-103

Protocol Name: A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and

**Activity Study of SYNT001 in Subjects with Chronic Pemphigus** 

(Vulgaris or Foliaceus)

IND Number: 132727

Study Drug: SYNT001

Protocol Version, Date: 2.0, 12-April-2017

**Clarification Letter Version: 2.0** 

Subjects: Infusion Reactions

**Concomitant Medications and Treatments** 

**Adverse Event Reporting** 

The purpose of this memo is to present planned revisions and required corrections in the protocol text resulting from requests for clarification from Investigators. Text regarding management of infusion reactions has been revised. Text regarding pre-medications has been added and text regarding adverse events that require reporting within 24 hours has been corrected. Deleted text is crossed through and new text is in italics.

This text will be formally revised in the next forthcoming protocol amendment. In the interim please provide this correspondence to your Institutional Review Board as per local policy.

#### Section 9.6.1 (page 63)

<u>Current Text:</u> Management of Grade 1 infusion reactions include decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen.

<u>Revised text:</u> Management of Grade 1 infusion reactions include *interrupting the infusion or* decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone <del>or</del> and acetaminophen, either alone or in combination, depending on the subject's signs and symptoms. If the infusion is interrupted

257 Park Ave S, 15<sup>th</sup> Floor, New York, New York, 10010

or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 (four) hours of SYNT001 preparation.

<u>Rationale:</u> Provides clarification for the management of a Grade 1 infusion reaction. Provides a maximum duration of infusion in accordance with the requirements for SYNT001 preparation and administration outlined in the pharmacy manual.

#### Figure 1 (page 64)

Title:

Current text: Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions

Revised Text: Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reactions

<u>Rationale</u>: To be consistent with prior section regarding management of a Grade 1 infusion reaction and with CTCAE v4.03 definition of a Grade 1 infusion reaction.

Last Box:

<u>Current text:</u> Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction

Revised Text: Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 preparation.

<u>Rationale</u>: Provision of a maximum duration of infusion in accordance with the requirements for SYNT001 preparation and administration as outlined in the pharmacy manual.

## Section 10 (page 69)

<u>Current text:</u> All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted.

Revised text: All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medications and treatments for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study (See Section 8.4.3). Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. Premedication is discouraged as prophylaxis against AEs or infusion reactions unless medically indicated from either past medical history, prior infusion reactions or AEs resulting from SYNT001 infusions.

Rationale: During recently conducted Site Initiation Visits for the Phase 1b studies of SYNT001, Syntimmune received questions about the possibility of infusion reactions with SYNT001. Indeed, infusion reactions are a common adverse effect of intravenous administration of monoclonal antibodies (mAb), even fully humanized mAbs. Infusion reactions are common with some FDA-approved mAbs, including anti-CD20 antibodies (Rituxan® [rituximab], Arzerra® [ofatumumab], Gazyva® [obinutumumab]), as well as with Cyramza® (ramucirumab) for gastric cancer, Darzelex® (daratumumab) for multiple myeloma, and Herceptin® (trastuzumab) for breast cancer. By contrast, infusion reactions are not reported in the package inserts for Soliris® (eculizumab) for paroxysmal nocturnal hemoglobinuria or Yervoy® (ipilimumab) for metastatic melanoma. Infusion reactions most commonly occur with the first infusion and are often related to the rate of protein infusion. For mAbs with frequent infusion reactions, it is typically recommended that pre-medications, such as corticosteroids, acetaminophen and an antihistamine, are administered prior to infusion, especially with the first infusion. For mAbs without associated infusion reactions or with uncommon or mild infusion reactions, premedications are not typically recommended and patients' signs and symptoms are managed individually.

While experience with SYNT001 is limited at this point, it is worth noting that there were no occurrences of infusion reactions in the recently completed healthy volunteer phase 1a single-

257 Park Ave S, 15th Floor, New York, New York, 10010

ascending dose study. In that study, infusions of SYNT001 were given over 1 hour at doses up to 30 mg/kg. No subject had their infusion interrupted or rate of infusion decreased. No subject received premedication prior to SYNT001 infusion.

While the phase 1a results for SYNT001 may not be indicative of what will be observed in future studies, Syntimmune does not currently believe that it is necessary or appropriate to administer pre-medications to patients who will be receiving SYNT001 at the same doses and same infusion rates as the healthy volunteers in the phase 1a study. Of course, sites must be prepared to manage infusion reactions from mild to severe during every infusion given in this study. Should an infusion reaction occur in any subject, their signs and symptoms should be managed as medically indicated, including the interruption of SYNT001 infusion or slowing of the rate of infusion. If frequent infusion reactions are observed in the phase 1b study, the issue of pre-medication will certainly be discussed with the investigators.

## Section 11.3.9.2 (page 76)

Cincoroly

<u>Current text:</u> "Any death, SAE, pregnancy, or unexpected (and severe) AE experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee)."

Revised text: "Any death, SAE, or pregnancy, or unexpected (and severe) AE experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee)."

<u>Rationale</u>: To clarify, adverse (severe) events that are not considered SAEs do not need to be reported within 24 hours but reported per section 11.3.6.

| Sincerely, | |
|---------------|------|
| PPD | |
| PPD | |
| Syntimmune, I | lnc. |

## SYNTIMMUNE

21-Sep-2017

**Protocol Number:** 

SYNT001-103

**Protocol Name:** 

A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and

**Activity Study of SYNT001 in Subjects with Chronic Pemphigus** 

(Vulgaris or Foliaceus)

**IND Number:** 

132727

**Study Drug:** 

SYNT001

**Protocol Version, Date:** 

2.0, 12-April-2017

Clarification Letter Version: 3.0

Subjects:

Inclusion Criteria

The purpose of this memo is to present a planned revision ahead of the next forthcoming protocol amendment. In the interim, please provide this correspondence to your Institutional Review Board as per local policy and request expedited review and approval.

#### Section 5.2 Inclusion Criteria #5 (page 35)

Current Text: Body mass index (BMI) 18.5 - 35.0 kg/m<sup>2</sup>

Revised text: Body mass index (BMI) 18.5 - 39.9 kg/m<sup>2</sup>

Rationale: Patients who may be otherwise eligible to participate in the study are excluded due to BMI. We would like to be able to offer these individuals the opportunity to participate.

Syntimmune, Inc.

257 Park Ave S, 15th Floor, New York, New York, 10010

## Syntimmune, Inc.

## **CLINICAL STUDY PROTOCOL**

## A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

Medical Monitor:

Wallace House

17-21 Maxwell Place Stirling, Scotland FK81JU

Mobile Phone: PPD

Office Phone: PPD

ext. PPD

 Original Protocol:
 18 January 2017

 Amendment 1.1:
 21 March 2017

 Amendment 2.0:
 12 April 2017

 Amendment 3.0:
 10 October 2017

#### **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

Page 403 of 979 Alexion Confidential

### **SPONSOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the Investigator, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| | 10-10-2017 |
|-----|-------------------|
| PPD | Date of Signature |
| | (DD Mm YYYY) |

## PROCEDURES IN CASE OF EMERGENCY

#### Serious Adverse Events

Any death or serious adverse event (SAE)\* occurring in a subject while receiving study drug or within 7 days of receiving study drug, even though the event may not appear to be study drug related, must be promptly reported (within 24 hours) by telephone or electronic communication to the sponsor (or designee).

## **Emergency Contact Information**

| For SAE reporting: | For any other questions or to contact the Medical Monitor: |
|---|---|
| Medpace Clinical Safety | PPD Mobile phone: PPD |
| Medpace SAE hotline: Telephone: PPD dial p or PPD | PPD Mobile phone: PPD |
| PPD dial P | Office phone: PPD ext. |
| Facsimile: PPD or PPD e-mail: PPD | PPD |
| | • |

## **SAE CRITERIA**

- \* A <u>serious adverse event</u> (SAE) is any untoward medical occurrence that at any dose results in any of the following outcomes, regardless of relationship to study drug (see <u>Section 11.3.1</u>, Serious Adverse Events for additional information):
  - Death
  - Life-threatening adverse drug event
  - Inpatient hospitalization or prolongation of existing hospitalization
  - A persistent or significant disability/ incapacity
  - A congenital anomaly/birth defect
  - An important medical event that may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

Syntimmune, Inc.


Amendment 3.0 Final 10October

## **INVESTIGATOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the sponsor, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonization Guideline for Good Clinical Practice (GCP), the Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

Nothing in this document is intended to limit the authority of a physician to provide emergency

| medical care under applicable regulations. | |
|---|---|
| Investigator Signature | Date of Signature<br>(DD Mm YYYY) |
| Name of Investigator (please print) | |

## 1 SYNOPSIS

| Study title | A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus) |
|---|---|
| Protocol number | SYNT001-103 |
| Number of study centers | Approximately 10 (US) |
| Clinical phase | Phase 1b |
| Study background | SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG immune complexes from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG containing immune complexes further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG immune complexes within and among compartments important in cellular immunity, it is further anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8+ and CD4+ T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG and IC that are involved in many autoimmune conditions and dismantle their ability to cause disease. SYNT001 targets mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP). While current treatments for certain autoimmune disorders including chronic steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are frequently associated with significant |
| | adverse effects, and delayed or non-durable responses. Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies are thought to play an important |

| | pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, leading to a significant decrease in total IgG, and thereby a corresponding decrease in the level of the pathogenic autoantibodies as well as the ICs to which they are associated, should lead to a decrease in the mucosal and cutaneous manifestations in subjects with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification. |
|---|---|
| Study rationale | This study is being conducted to further evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers. |
| Study objectives | Primary objective |
| | To evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus) |
| | Secondary objectives |
| | To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels |
| | To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers: |
| | <ul> <li>Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM</li> <li>Albumin</li> </ul> |
| | • To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers: |
| | <ul> <li>Serum anti-desmoglein (Dsg) (1 and 3) antibody levels</li> </ul> |
| | o Pemphigus Disease Area Index (PDAI) |
| | To assess immunogenicity (anti-SYNT001 antibodies) |
| | Exploratory objectives |
| | To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including: |
| | <ul> <li>Serum anti-epithelial cell antibody (AECA) levels by indirect<br/>immunofluorescence</li> </ul> |
| | Circulating immune complexes (CIC) |
| | o Complement component 3 (C3) |
| | <ul> <li>Exploratory biomarkers (FCGR2A (single nucleotide polymorphism-<br/>SNP), RNAseq, urine IgG)</li> </ul> |

| 0 | Immune phenotyping by flow cytometry for CD3 <sup>+</sup> CD4 <sup>+</sup> T, |
|---|---|
| | CD3 <sup>+</sup> CD8 <sup>+</sup> T, monocytes, NK cells and B cells |

- SYNT001 levels in skin biopsies (optional)
- Exploratory biomarkers to investigate immune response associated with pemphigus
- To characterize corticosteroid use during the study

#### Study design

Phase 1b, multicenter, open-label, safety, tolerability, and activity study

#### Methodology

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of subjects | Dose |
|--------|-----------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs, and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All safety data and any available and relevant PD data through Day 42 (2 weeks after the last subject's last dose in Cohort 1) will be reviewed by a dose escalation committee before Cohort 2 is initiated. Escalation to Cohort 2 will proceed if there are no concerning safety signals and the review of available and relevant PD data supports advancing to a higher dose. The dose for Cohort 2 will be finalized after review of the safety and PD data, but will not exceed 30 mg/kg. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule as Cohort 1.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the

6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33. On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84 and 112. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made. Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42 and 56 for safety assessments, study drug dosing, sample collections, and other study procedures. Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management. See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, adverse event (AE) assessments, concomitant medication assessments, and electrocardiograms (ECG). Approximately 16; two cohorts of 8 subjects each. An additional cohort of up to Number of subjects 8 subjects may be enrolled. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects with pemphigus foliaceus may be enrolled. Diagnosis and main **Inclusion criteria:** entry criteria Subjects must meet the following criteria to be included: 1. Willing and able to read, understand and sign an informed consent form; 2. Male or female  $\geq$  18 years of age at the time of screening; 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria: a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions): b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal; c. History of at least one positive tissue-based test (e.g., biopsy, direct immunofluorescence [DIF]) 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:

- a. If treated with rituximab or other anti-CD20 antibodies, last dose
   12 months prior to screening;
- b. If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
- c. If being treated with corticosteroids, must be ≤ 1mg/kg/day of prednisone or equivalent and stable (< 10% change in dose) for 2 weeks prior to screening;
- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 39.0 \text{ kg/m}^2$ ;
- 6. Has a negative pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intra-uterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through the final study visit.

#### **Exclusion criteria:**

Subjects meeting any of the following criteria are to be excluded:

- 1. Subject unable or unwilling to comply with the protocol;
- 2. Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG use within 60 days of screening;
- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;

| | <ol> <li>Any exposure to an investigational drug or device within the 30 days prior to screening</li> <li>Plasmapheresis or immunoadsorption within 60 days of screening</li> <li>Cellular therapy, including CAR-T, at any time prior to screening</li> <li>Use of any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of screening</li> <li>Serum total IgG &lt; 600 mg/dL;</li> <li>Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (e.g., a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results);</li> <li>Any vaccination within 2 weeks of screening</li> </ol> |
|---|---|
| Study drug, dosage, | SYNT001 |
| and administration | <b>Doses:</b> 10 mg/kg and 30 mg/kg. A third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive. |
| | SYNT001 is provided as a liquid at a nominal concentration of 50 mg/mL. SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for infusion. |
| | Route of administration: IV in 250 mL over 1 hour |
| Control, dose, and route of administration | Not applicable |
| Duration of subject participation and duration of study | Up to 126 days (18 weeks): Screening of up to 2 weeks (14 days); Treatment period of 8 weeks (56 days); Follow-up period of 8 weeks (56 days) |

## Prohibited Concomitant treatments

All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. Premedication is discouraged as prophylaxis against AEs or infusion reactions unless medically indicated from either past medical history, prior infusion reactions or AEs resulting from SYNT001 infusions.

Use of the following medications will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations through Day 56. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator.

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

#### Safety assessments

Safety assessments include AEs, serious adverse events (SAEs), PEs, vital sign measurements, clinical safety laboratory evaluations, ECGs, and reasons for treatment discontinuations due to toxicity. Safety assessments will be performed at specified time points and prior to discharge from the clinic. Vital sign measurements, including blood pressure, pulse rate, respiratory rate, and temperature will be monitored throughout the study. Pulse oximetry will be monitored during the study drug infusion and for 2 hours following the end of the infusion.

| | The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03) will be used for grading clinical and laboratory AEs. The AE reporting period for a subject enrolled in the study begins when the subject provides informed consent and is continued through the last study visit. All AEs that occur in the enrolled subjects during the AE reporting period must be recorded, regardless of the relationship of the AE to study drug. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug should also be recorded. |
|---|---|
| Dose-escalation rules | Dose escalation decisions will be made by a Dose Escalation Committee (DEC) and will be based on safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities, AEs, SAEs, and total IgG levels. Dose-limiting toxicity (DLT) will be defined generally as severe (Grade 3) AEs occurring in ≥ 2 subjects that are determined to be clinically significant and considered related to study drug. If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. If the dose-escalation stopping rule is met during Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics data will be reviewed and the cohort may resume (if applicable) or a new cohort may be added, at a dose at least 50% lower than the |
| | 10 mg/kg dose. If the stopping rule is not met in Cohort 1 (10 mg/kg), dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met for the first time during Cohort 2, all safety data and all available pharmacodynamics data will be reviewed and the cohort may resume (if applicable) or a new cohort may be added at a dose at least 30% lower than the Cohort 2 dose. If the stopping rule is not met in Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data. |
| Study stopping rule | If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, any further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the next appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects. |
| Individual stopping rule | Dosing for any individual subject will be discontinued (i.e., further treatment with the study drug will not be given) if the subject experiences any study drug- |

| | related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject will be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in dose(s) of antipemphigus medication(s) for the management of pemphigus. |
|---|---|
| Pharmacokinetics | The PK of SYNT001 will be evaluated following the first and last (fifth) doses of SYNT001. |
| | Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. Study drug concentration will be used to calculate the following PK parameters: $t_{1/2}$ , $C_{max}$ , $T_{max}$ , $AUC_{0-24}$ , and $AUC_{0-\infty}$ . |
| Pharmacodynamics/<br>Activity | PD samples will be collected for analysis of IgG (serial assessment of IgG levels to identify C <sub>min</sub> , T <sub>min</sub> ); IgG1-4 subtype levels; IgA levels; IgM levels; albumin levels; anti-Dsg (1 and 3) antibody levels; serum AECA by direct immunofluorescence; CIC; C3; exploratory biomarkers ( <i>FCGR2A</i> SNP, RNAseq, urine IgG, CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T, monocytes, NK cells and B cells), and additional exploratory analyses to investigate immune response associated with pemphigus. |
| Immunogenicity | Samples will be collected for immunogenicity analyses on Days 0 (pre-dose), 14, 28, 56, 84 and 112. |
| Skin biopsy | Optional skin biopsy samples from lesional or non-lesional skin will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33, 56 and 84 to analyze SYNT001 levels. |
| Photography | Photographs of active lesions will be taken at Day 0. Follow-up photographs of the same areas will be taken on Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. |
| Statistical methods | Sample size consideration |
| | Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives. |
| | Data presentations/Descriptive statistics |
| | Three populations will be employed in the analysis of study data. |

- The intent-to-treat (ITT) population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population.
- The PK population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters.
- The PD population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the PK and ITT populations, where appropriate.

#### Criteria for evaluation

| Objective | Endpoint |
|---|---|
| Primary | - |
| Safety and tolerability of 5 once-<br>weekly IV infusions of SYNT001 to<br>subjects with pemphigus vulgaris or<br>foliaceus | AEs and clinical (safety) laboratory tests |
| Secondary | |
| PK of SYNT001 following a 1-hour IV infusion | PK parameters: $t_{1/2}$ , $C_{max}$ , $T_{max}$ , $AUC_{0-24}$ , and $AUC_{0-\infty}$ . |
| Effect of 5 once-weekly IV doses of SYNT001 on: • Total IgG (IgG1-4), IgA, IgM, and albumin • Serum anti-Dsg (1 and 3) antibodies | Changes in levels of IgG, IgG subtypes (IgG1-4), IgA, IgM, albumin, serum anti-Dsg (1 and 3) antibodies |
| Assess immunogenicity | Anti-SYNT001 antibodies |
| Disease Activity | PDAI Scores |
| Exploratory | |
| Effect of 5 once-weekly IV doses of SYNT001 on biomarkers including: • CIC • C3 • Serum anti-epithelial cell antibody (AECA) levels • Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG) • Immune phenotyping by flow cytometry | Changes in CIC; C3; AECA levels by indirect immunofluorescence; <i>FCGR2A</i> SNP; RNAseq; urine IgG, CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T, monocytes, NK cells and B cells; urine IgG levels; changes in blood transcriptome |

| Exploratory biomarkers to<br>investigate immune response<br>associated with pemphigus | |
|---|---|
| Concomitant Treatment | Corticosteroid use during the study |
| SYNT001 levels in skin biopsies | Measures of SYNT001 levels in skin biopsies |

Treatment-emergent AEs (TEAEs) will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, or treatment discontinuation will be listed by subject, and cohort using SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken, and outcome.

Laboratory results will be summarized by time point and cohort. The incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the central laboratory. Vital sign measurements will be summarized by cohort at each scheduled time point using descriptive statistics.

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and area under the curve (AUC). PK parameters will be determined using non-compartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

PD results will be summarized by cohort. Descriptive statistics of PD parameters for SYNT001 will include mean, SD, CV, median, minimum, and maximum.

Immunogenicity results will be summarized by cohort. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

**Table 1:** Study Assessments

| | Screening | | Treatment Period | | | | | | | F | ollow-Up | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timepoint (Study Day) | -14 to -1 | 0 | 1<br>(±1<br>hr) | 2<br>(± 2<br>hr) | 5 <sup>p</sup><br>(±4<br>hr) | 7<br>(±6<br>hr) | 12 <sup>p</sup><br>(±6<br>hr) | 14<br>(±6<br>hr) | 19 <sup>p</sup><br>(±6<br>hr) | 21<br>(±6<br>hr) | 28<br>(±6<br>hr) | 29<br>(±1<br>hr) | 30<br>(±2<br>hr) | 33<br>(±4<br>hr) | 42<br>(±3<br>days) | 56<br>(±5<br>days) | 84<br>(±5<br>days) | 112<br>(±5 days) or ET<br>Visit |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Demographics/Medical History | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>a</sup> | X | X | | | | X | | X | | X | X | | | | X | X | X | X |
| Vital Signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse Oximetry <sup>c</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Clinical Safety Labs <sup>d</sup> | X | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis & HIV Screen | X | | | | | | | | | | | | | | | | | |
| 12-Lead ECG <sup>f</sup> | X | X | | | | | X | | | | X | | | | | X | | |
| Tetanus & VZV antibodies | | X | | | | | | | | | | | | | | X | X | X |
| PDAI Score | | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| PK Sampling <sup>h</sup> | | X | X | X | X | | | | | | X | X | X | X | | | | |
| Immunogenicity <sup>i</sup> | | X | | | | | | X | | | X | | | | | X | X | X |
| Study Drug Administration <sup>j</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4) <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>q</sup> |
| CIC | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Anti-Dsg (1 & 3) antibody titer | X | X | | | | X | | X | | | | | | X | | X | X | X |
| C3 and AECA <sup>1</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| FCGR2A <sup>m</sup> by buccal swab | | X | | | | | | | | | | | | | | | | |
| RNAseq <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| Urine IgG <sup>m</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| Immune phenotyping <sup>n</sup> | | X | | | | | | | | | X | | | | | X | | |
| Pemphigus immune response biomarkers | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Optional Skin Biopsy | | X | X | X | | | | X | | | | | | X | | X | X | |
| Photography <sup>o</sup> | | X | | | | | | | | | | | | X | | X | X | X |
| Adverse Events | | | | | To be | e collec | ted fron | n the da | te that i | the ICF | is signe | ed throu | igh the i | last study | visit | | | |
| Concomitant Medications | | | | | To be | e collec | ted fron | n within | 14 day | s prior | to Day | 0 throu | gh the i | last study | visit | | | |

ECG = electrocardiogram; ET= Early Termination; HIV = human immunodeficiency virus; ICF = informed consent form; PD = pharmacodynamic; PK = pharmacokinetic; VZV = varicella-zoster virus

Syntimmune, Inc.


Amendment 3.0 Final 10 October 2017

- a: Complete PE, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.
- b: **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. On Days 0, 7, 14, 21, and 28 vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- c: **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d: Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 6.7 for a complete list). Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 112.
- e: **Pregnancy test:** To be performed at time of screening and prior to first dose of SYNT001 on Day 0 and on Days 56 and 112 (urine or serum test is acceptable, however, positive urine tests must be confirmed with serum testing.)
- f: Digital 12-lead **ECG** to be obtained after 5 minutes of rest in the supine position and in triplicate at least 1-2 minutes apart (see Section 6.6 for additional information). On Days 0 and 28 to be obtained 5 minutes after the completion of infusion. Day 12 ECG will be collected only if the visit is conducted at the study site.
- g: **Serology**: Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 84; if still below the baseline value (or level of detection), the subject will be re-tested at Day 112. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112, will be referred to their primary care physician for further management. See Section 6.7.3 for additional information.
- h: **PK:** Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. See Section 6.7.4 for additional information.
- i: Immunogenicity: Blood samples will be collected pre-dose when collected on dosing days. Samples will be collected on Days 0, 14, 28, 56, 84 and 112. See Section 6.7.6 for additional information.
- j: Prior to **study drug infusion**, SYNT001 drug product is to be diluted in Dextrose 5% in Water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour using a 0.2-micron, inline filter. See Section 9 for additional information.
- k: Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, and IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 6.7.5 for additional information
- 1: Exploratory PD samples (C3 and AECA): collected pre-dose when collected on dosing days. See Section 6.7.5 for complete information.
- m: Buccal samples to be collected and stored; pending review of clinical and pharmacodynamics assessments
- n: Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- o: Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- p: Visit Days 5, 12 and 19 may be conducted via at-home nursing in lieu of a subject visit to the study site.
- q: Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

Table 2: Timing Window Allowances for PK/PD Sampling, ECG, and Vital Sign Measurements

| Pharmacokinetic and Pharmacodynamic Sampling | |
|------------------------------------------------|-------------------------|
| Timepoint | <b>Tolerance Window</b> |
| 0 hour | −240 min to 0 hour |
| 5 minutes post end-of-infusion | ± 5 minutes |
| 2, 4, & 6 hours post end-of-infusion | ± 15 minutes |
| 24 hours post end-of-infusion | $\pm$ 60 minutes |
| 48 hours post end-of-infusion | ± 120 minutes |
| ECG | |
| Timepoint | <b>Tolerance Window</b> |
| 5 minutes post end-of-infusion | $\pm 10$ minutes |
| Vital Signs <sup>a</sup> | |
| Timepoint | <b>Tolerance Window</b> |
| 0 hour | −240 min to 0 hour |
| 15, 30, and 45 minutes after start of infusion | ± 5 minutes |
| 60 minutes after start of infusion | ± 10 minutes |
| 30, 60 and 120 minutes post end-of-infusion | $\pm 10$ minutes |

a: Vital signs to include blood pressure, pulse rate, respiratory rate, oral temperature, and pulse oximetry.

## TABLE OF CONTENTS

| PROCE | DURES IN CASE OF EMERGENCY | 3 |
|--------|---------------------------------------------|----|
| INVEST | ΓΙGATOR SIGNATURE | 4 |
| 1 SY | YNOPSIS | 5 |
| LIST O | F ABBREVIATIONS | 24 |
| 2 BA | ACKGROUND AND RATIONALE | 26 |
| 2.1 | Study Rationale | 27 |
| 2.2 | Selection of Doses in this Study | |
| 2.3 | Compliance Statement | |
| 3 ST | TUDY OBJECTIVES | 29 |
| 3.1 | Primary Objective | 29 |
| 3.2 | Secondary Objectives | 29 |
| 3.3 | Exploratory Objectives | 29 |
| 4 ST | TUDY DESIGN | 30 |
| 4.1 | Study Sites | 30 |
| 4.2 | Study Endpoints | 30 |
| 4.3 | Overview of Study Design | 31 |
| 4.4 | Randomization and Blinding | 33 |
| 5 ST | TUDY POPULATION | 34 |
| 5.1 | Target Population | 34 |
| 5.2 | Inclusion Criteria | 34 |
| 5.3 | Exclusion Criteria | 35 |
| 6 ST | TUDY PROCEDURES | |
| 6.1 | Informed Consent | |
| 6.2 | Demographics and Medical History | 37 |
| 6.3 | Physical Examination | |
| 6.4 | Pemphigus Disease Area Index (PDAI) Scoring | 37 |
| 6.5 | Vital Sign Measurements | |
| 6.6 | 12-Lead Electrocardiogram (ECG) | |
| 6.7 | Clinical Laboratory Measurements | |
| | 6.7.1 Pregnancy Testing | |
| | 6.7.2 Virology | 40 |

| | | 6.7.3 | Serum Tetanus Antibody and Varicella-Zoster Virus Antibody | Testing40 |
|---|---|---|---|---|
| | | 6.7.4 | Pharmacokinetics (PK) Sampling | 41 |
| | | 6.7.5 | Pharmacodynamic Sampling | 41 |
| | | 6.7.6 | Immunogenicity Testing | 42 |
| | 6.8 | Study | Drug Administration | 43 |
| | 6.9 | Prior | and Concomitant Medications | 43 |
| | 6.10 | Adve | rse Event Assessments | 43 |
| | 6.11 | Photo | graphs | 44 |
| | 6.12 | Skin l | Biopsy | 44 |
| 7 | ST | UDY AS | SSESSMENTS | 45 |
| | 7.1 | Scree | ning Period: Day -14 to Day -1 | 45 |
| | 7.2 | Enrol | lment and First Treatment: Day 0 | 45 |
| | 7.3 | | w-up: Day 1 | |
| | 7.4 | Follo | w-up: Day 2 | 47 |
| | 7.5 | Follo | w-up: Day 5 | 48 |
| | 7.6 | Treati | ment Day 7 (Dose 2) | 48 |
| | 7.7 | Dose | 2 Follow-up Day 12 | 49 |
| | 7.8 | Treati | ment Day 14 (Dose 3) | 49 |
| | 7.9 | Dose | 3 Follow-up Day 19 | 51 |
| | 7.10 | Treati | ment Day 21 (Dose 4) | 51 |
| | 7.11 | Treati | ment Day 28 (Dose 5) | 52 |
| | 7.12 | Follo | w-up Day 29 | 53 |
| | 7.13 | Follo | w-up Day 30 | 54 |
| | 7.14 | Follo | w-up Day 33 | 54 |
| | 7.15 | Follo | w-up Day 42 | 55 |
| | 7.16 | Follo | w-up Day 56 | 55 |
| | 7.17 | Follo | w-up Day 84 | 56 |
| | 7.18 | Follo | w-up Day 112 (End-of-Study) or Early Termination Visit | 57 |
| 8 | RE | MOVIN | IG SUBJECTS FROM STUDY | 58 |
| | 8.1 | Subje | ct Withdrawal | 58 |
| | 8.2 | Study | Discontinuation | 59 |
| | 8.3 | Repla | cements | 59 |
| | 8.4 | Stopp | ing Rule | 59 |
| | | 8.4.1 | Dose-Escalation Stopping Rule | |
| | | 8.4.2 | Study Stopping Rule | |
| | | 8.4.3 | Individual Stopping Rule | 60 |

| 9 | ST | UDY DR | UG | 61 |
|---|---|---|---|---|
| | 9.1 | SYNT | 001 | 61 |
| | 9.2 | | t Dosing | |
| | 9.3 | | g of Dosing | |
| | 9.4 | | y of Investigational Products | |
| | 9.5 | | gational Product Retention at Study Site | |
| | 9.6 | | ngs and Precautions | |
| | | 9.6.1 | Infusion Reaction | |
| | | 9.6.2 | Potential Immune Effects | 67 |
| 10 | CC | NCOMI | TANT MEDICATION AND TREATMENT | 69 |
| 11 | SA | FETY | | 71 |
| | 11.1 | Safety | Parameters | 71 |
| | 11.2 | Advers | se Event Definition | 71 |
| | 11.3 | Evalua | ting Adverse Events | 72 |
| | | 11.3.1 | Serious Adverse Events | 72 |
| | | 11.3.2 | Overdose | 73 |
| | | 11.3.3 | Non-Serious Adverse Events | 73 |
| | | 11.3.4 | Protocol-Related Adverse Events | 73 |
| | | 11.3.5 | Assessment of Causality | 73 |
| | | 11.3.6 | Recording Adverse Events | 74 |
| | | 11.3.7 | Planned Hospitalization | 74 |
| | | 11.3.8 | Reporting Pregnancies | 75 |
| | | 11.3.9 | Serious Adverse Event Reporting. | 75 |
| | | 11.3.9.1 | Governing Regulatory Requirements | 75 |
| | | 11.3.9.2 | Time Frame for Reporting | 76 |
| | | 11.3.9.3 | Information to be Provided by the Investigator | 77 |
| | | 11.3.10 | Regulatory Reporting | 78 |
| | | 11.3.11 | Follow-up Information on a Serious Adverse Event (SAE) | 79 |
| | 11.4 | Other | Safety Considerations | 79 |
| | | 11.4.1 | Laboratory Data | 79 |
| | | 11.4.2 | Medication Errors | 79 |
| | | 11.4.3 | Follow-Up of Adverse Events | 79 |
| | 11.5 | Safety | Monitoring for Dose Escalation | 79 |
| 12 | ST | ATISTIC | AL CONSIDERATIONS | 81 |
| | 12.1 | Genera | al Design | 81 |
| | 12.2 | | e Size Justification | |
| | 12.3 | Statist | ical Considerations | 81 |

| | | 12.3.1 Study Populations | 81 |
|---|---|---|---|
| | | 12.3.2 Subject Accountability, Demographics, and Baseline Characterists | ics 82 |
| | | 12.3.3 Concomitant Medications | 82 |
| | 12.4 | Planned PK Analysis | 82 |
| | 12.5 | Safety Data | 83 |
| | 12.6 | Pharmacodynamic/Activity Data | 83 |
| | 12.7 | Immunogenicity Data | 83 |
| | 12.8 | Interim Analysis | 84 |
| 13 | DA | ATA QUALITY ASSURANCE | 85 |
| 14 | ST | UDY ADMINISTRATION | 86 |
| | 14.1 | Study Administrative Structure | 86 |
| | 14.2 | Ethical Conduct of the Study | 86 |
| | 14.3 | Informed Consent (ICF) | 86 |
| | 14.4 | Institutional Review Board | 87 |
| | 14.5 | Dose Escalation Committee | 87 |
| | 14.6 | Future Use of Subject Samples | 88 |
| 15 | CC | ONDITIONS FOR MODIFYING THE PROTOCOL | 89 |
| 16 | CC | ONDITIONS FOR TERMINATING THE STUDY | 90 |
| 17 | ST | UDY DOCUMENTATION, CRFS, AND RECORD KEEPING | 91 |
| | 17.1 | Investigator's Files and Retention of Documents | 91 |
| | 17.2 | Source Documents and Background Data | 91 |
| | 17.3 | Audits and Inspections | 92 |
| | 17.4 | Electronic Case Report Forms | 93 |
| 18 | MO | ONITORING THE STUDY | 94 |
| 19 | CC | ONFIDENTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECORDS | S95 |
| 20 | PU | BLICATION OF DATA AND PROTECTION OF TRADE SECRETS | 96 |
| 2 1 | DE | FEDENCES | 07 |

| T | IST | OF | T 1 | RI | FS |
|---|------|----|-----|------|-------|
| | 1101 | vi | 1 / | . DI | 1 1/1 |

| Table 1: | Study Assessments | 16 |
|---|---|---|
| Table 2: | Timing Window Allowances for PK/PD Sampling, ECG, and Vita | ıl Sign |
| | Measurements | 18 |
| Table 3: | Clinical Laboratory Panels | 39 |
| Table 4: Ph | narmacodynamic/ Activity Assessments | |
| Table 5: | Grading and Management of Allergic or Infusion-Related Reaction | ns 66 |
| Table 6: | Study Administrative Structure | 86 |
| LIST OF I | | |
| • | Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reaction | |
| Figure 2: N | Management of Severe (Grade 3 or higher) Infusion Reactions | 65 |
| LIST OF A | APPENDICES | |
| Appendix A | A: NCI CTCAE, Version 4.03 | 99 |
| Appendix I | R. Pemphigus Disease Area Index | 100 |

#### LIST OF ABBREVIATIONS

ADA Anti-drug antibodies

AE Adverse event

AECA Anti-epithelial cell antibody
ALT Alanine aminotransferase
ANA Antinuclear antibody
AST Aspartate aminotransferase
ATC Anatomical therapeutic chemical

AUC<sub>0.24</sub> Area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose

 $AUC_{0\text{--}\infty} \qquad \qquad \text{Area under the plasma concentration-time curve from pre-dose (time 0) to infinity}$ 

BLQ Below the limit of quantification

BMI Body mass index
BUN Blood urea nitrogen

CAR-T Chimeric antigen receptor and T-cell

CFR Code of Federal Regulations
C3 Complement component 3
CBC Complete blood count

CIC Circulating immune complexes

CIDP Chronic inflammatory demyelinating polyneuropathy

C<sub>max</sub> Maximum plasma concentration determined directly from the concentration-time profile

CRO Contract research organization

CV Coefficient of variation

CVID Common variable immune deficiency

DEC Dose escalation committee
D5W Dextrose 5% in Water
DIF Direct immunofluorescence
DNA Deoxyribonucleic acid
ECG Electrocardiogram

eCRF Electronic case report form
ESR Erythrocyte sedimentation rate
FcGR2a Fc Gamma R2a receptor
FcRn Neonatal Fc receptor

FDA Food and Drug Administration

GCP Good Clinical Practice

GI Gastrointestinal
HBV Hepatitis B virus
HCV Hepatitis C virus

HIPAA Health Insurance Portability and Accountability Act

HIV Human immunodeficiency virus

IB Investigator's brochure IC Immune complex

ICF Informed consent form

ICH International Conference on Harmonization

IgA Immunoglobulin A
IgG Immunoglobulin G
IgG1-4 Immunoglobulin G1-G4
IgM Immunoglobulin M
IL-12 Interleukin 12

IND Investigational new drug
IRB Institutional review board

ITT Intent-to-treat
IUD Intrauterine devices

IV Intravenous

IVIG Intravenous immunoglobulin

MedDRA Medical Dictionary for Regulatory Activities

NHL Non-Hodgkin lymphoma
PD Pharmacodynamics
PE Physical examination
PK Pharmacokinetic
RBC Red blood cells
RNAseq RNA sequencing

QTcF Corrected QT interval using Fridericia's formula

SAE Serious adverse event SAP Statistical analysis plan SAS Statistical Analysis System

SD Standard deviation

SNP Single nucleotide polymorphism

SOC System Organ Class

SOP Standard operating procedures

SYNT001 A humanized, affinity matured IgG4-kappa monoclonal antibody

t<sub>1/2</sub> Half-life

TEAE Treatment-emergent adverse event

T<sub>max</sub> Observed time to reach peak plasma concentration

TNF Tumor necrosis factor ULN Upper limit of normal

UNS Unscheduled

VZV Varicella-zoster virus

WAIHA Warm antibody autoimmune hemolytic anemia

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

#### 2 BACKGROUND AND RATIONALE

SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks IgG and IgG immune complex (IC) interactions with the neonatal Fc receptor (FcRn) and thereby the major functions of FcRn in protecting IgG and IgG ICs from degradation and their role in downstream signaling events. Specific and high affinity blockade of FcRn with SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-antigen IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG-containing ICs further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen-presenting cells will result in inhibition of IC-stimulated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG ICs within and among compartments important in cellular immunity, it is anticipated that SYNT001 will block antigen processing and presentation of antigens contained within IC that otherwise lead to CD8<sup>+</sup> and CD4<sup>+</sup> T cell activation. Thus, SYNT001 will specifically target immune functions associated with IgG that are involved in certain autoimmune conditions and dismantle their ability to cause disease.

SYNT001 targets key mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm antibody autoimmune hemolytic anemia (WAIHA), pemphigus, and chronic inflammatory demyelinating polyneuropathy (CIDP).

While current treatments for certain autoimmune disorders, including high-dose steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they are associated with significant adverse effects, as well as delayed or non-durable responses.

Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies have been shown to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, which significantly decreases total IgG, including a corresponding decrease in the level of the pathogenic autoantibodies and the ICs to which they are associated, may lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for further sustained disease modification.

## 2.1 Study Rationale

This study is being conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers.

## 2.2 Selection of Doses in this Study

The planned dose levels of SYNT001 for this Phase 1b safety and proof-of-concept study of 10 mg/kg and 30 mg/kg were selected from careful review of the safety, tolerability, and PD effect on total IgG levels after single and repeat dosing of SYNT001 in non-human primates (NHPs), as well as the safety, tolerability, and PD effect on total IgG levels after single ascending doses of SYNT001 in healthy volunteers. In addition, further consideration was given to the desired level of FcRn blockade to achieve suppression of IgG to a range that has been previously correlated with disease remission. Further, we considered the potential effects of inhibiting FcRn function as they relate to immune complex associated innate and adaptive immunity in choosing these dose levels based upon exploratory studies of a single ascending dose of SYNT001 in healthy volunteers. From the NHP studies, single doses of SYNT001 produced a dose-dependent decrease in total IgG and a further decrease was seen with repeated weekly doses up to a maximum 70% reduction at 100 mg/kg. This magnitude of total IgG reduction is approaching the expected maximal effect of 100% inhibition of FcRn function based on murine studies also performed by Syntimmune and others (Nixon et al., 2015; Roopenian et al., 2003). In the recently completed Phase 1a trial with SYNT001 in healthy volunteers a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the NHP studies further reductions are expected following multiple dosing. A comparable decrease in pathogenic autoantibodies is also anticipated.

In the NHP studies, relevant adverse effects, mild-to-moderate infusion reactions, were observed only after the third weekly IV administration, concurrent with the development of anti-SYNT001 antibodies. In the recently completed Phase 1a healthy male volunteer study, the doses of SYNT001 up to and including 30 mg/kg have been well tolerated. There were no dose limiting toxicities, serious adverse events, or any other safety concerns identified. No AEs were observed in the 1 and 3 mg/kg dose cohorts. A single Grade 2 AE was observed; a headache in the 10 mg/kg cohort. Other subjects had mild (Grade 1) AEs at 10 mg/kg. In Cohort 4 (30 mg/kg), 5 subjects received SYNT001. All five subjects experienced AEs; all were mild (Grade 1), transient and resolved spontaneously without intervention. Therefore, it is anticipated that the doses selected for this study should be well tolerated and have clinically relevant PD effects in patients with chronic pemphigus (vulgaris or foliaceus). For a summary of findings from the

single dose, clinical study in healthy subjects and further details on the nonclinical findings, please refer to the SYNT001 Investigator's Brochure.

## 2.3 Compliance Statement

This study will be conducted in compliance with Good Clinical Practice (GCP), including the International Conference on Harmonisation (ICH) Guidelines and FDA regulations, consistent with the principles outlined in the Declaration of Helsinki. In addition, the Investigator agrees to adhere to all applicable local laws and regulatory requirements relevant to the use of new therapeutic agents.

The study will be conducted in compliance with the protocol. The appropriate Institutional Review Boards (IRBs) must approve the protocol, any amendments, and the subject informed consent form (ICF) prior to implementation.

Freely given written informed consent must be obtained from every subject prior to participation in this clinical trial. As part of this procedure, the Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or AEs that may occur. The study subject should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The Investigator or designee will provide the Sponsor with a copy of the IRB-approved informed consent form prior to the start of the study. The rights, safety, and well-being of participating subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (e.g., loss of medical licensure, debarment).

#### 3 STUDY OBJECTIVES

## 3.1 Primary Objective

The primary objective of this study is to evaluate the safety and tolerability of 5 once-weekly IV infusions of SYNT001 at different dose levels in subjects with chronic pemphigus (vulgaris or foliaceus).

## 3.2 Secondary Objectives

The secondary objectives of this study are as follow:

- To determine the PK of SYNT001 following 5 once-weekly 1-hour IV infusions at different dose levels
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following PD biomarkers:
  - o Immunoglobulins: IgG, IgG subtypes (IgG1-4), IgA, IgM
  - o Albumin
- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following disease activity markers:
  - o Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
  - o Pemphigus Disease Area Index (PDAI)
- To assess immunogenicity (anti-SYNT001 antibodies)

### 3.3 Exploratory Objectives

The exploratory objectives of this study are as follow:

- To assess the effect of 5 once-weekly doses of SYNT001 at different dose levels on the following biomarkers, including:
  - o Serum anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence
  - o Circulating immune complexes (CIC)
  - o Complement component 3 (C3)
  - Exploratory biomarkers (FCGR2A single nucleotide polymorphism-SNP, RNAseq, urine IgG)
  - Immune phenotyping by flow cytometry for CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
  - o SYNT001 levels in skin biopsies (optional)
  - o Exploratory biomarkers to investigate immune response associated with pemphigus
- To characterize corticosteroid use during the study
#### 4 STUDY DESIGN

#### 4.1 Study Sites

This study will be conducted at approximately 10 sites in the United States (US).

#### 4.2 Study Endpoints

**Primary Outcome Measures:** Assessment of safety data (adverse events [AEs], serious adverse events [SAEs], vital sign measurements, ECGs and clinical laboratory tests) will be the primary safety measure.

#### **Secondary Outcome Measures**

#### Pharmacokinetics:

Half-life (t<sub>1/2</sub>), maximum plasma concentration determined directly from the concentration-time profile (C<sub>max</sub>), observed time to reach peak plasma concentration (T<sub>max</sub>), area under the plasma concentration-time curve from pre-dose (time 0) to 24 hours post-dose (AUC<sub>0-24</sub>), and area under the plasma concentration-time curve from pre-dose (time 0) to infinity (AUC<sub>0-∞</sub>)

#### PD Biomarkers:

- Ig Assessments: Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o Serial assessments of total IgG and IgG subtypes (IgG1-4)
  - o IgA levels
  - o IgM levels
- Albumin levels

#### Disease activity markers:

- Serum anti-desmoglein (Dsg) (1 and 3) antibody levels
- Pemphigus Disease Area Index (PDAI) scores

#### Immunogenicity:

• Anti-SYNT001 antibodies

#### **Exploratory Outcome Measures**

Biomarkers, including:

- CIC
- C3
- Serum AECA levels
- Exploratory biomarkers (FCGR2A SNP, RNAseq, urine IgG)

- Immune phenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells
- SYNT001 levels in skin biopsies (optional)
- Exploratory biomarkers to investigate immune response associated with pemphigus

#### **Concomitant Treatments**

Corticosteroid use

Further details on the statistical and analytical plan for these endpoints are available in Section 12, Statistical Considerations.

### 4.3 Overview of Study Design

This will be a multicenter, open-label study to assess the safety, tolerability, activity, PK, PD, and immunogenicity of 5 once-weekly IV infusions of SYNT001 to subjects with chronic pemphigus (vulgaris or foliaceus).

Planned doses of SYNT001 to be studied are 10 mg/kg and up to 30 mg/kg. Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 10 mg/kg or up to 30 mg/kg. Based on review of safety, PD, and clinical outcomes of the first cohort, the dose for the second cohort may be adjusted, but with a maximum dose of 30 mg/kg. Based on review of safety, PD and clinical outcomes from these 2 cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort | No. of<br>Subjects | Dose |
|--------|--------------------|------------------|
| 1 | 8 | SYNT001 10 mg/kg |
| 2 | 8 | SYNT001 30 mg/kg |

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. This evaluation will include a review of AE/SAE reports, vital sign assessments, physical examinations, ECGs and clinical laboratory testing. The seriousness, severity, and relatedness of AEs/SAEs will also be considered in the safety evaluation. Safety data will be reviewed on a continuous basis throughout the study. All data through Day 42

(2 weeks after the last subject's last dose in Cohort 1) will be reviewed before Cohort 2 is initiated. Cohort 2 and Cohort 3, if added, will be dosed per the same schedule.

Safety evaluations will be conducted by a dose escalation committee (DEC). The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions. Dosing and dose escalation will proceed if the DEC has determined that it would be safe and appropriate to do so. In addition, over the course of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects.

On days where study drug is administered, vital sign and pulse oximetry measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.

On Days 0 and 28, PK blood samples will be collected prior to infusion start and then over the subsequent 48 hours. Subjects will remain at the clinic through the 6-hour PK sample collection and will return to the clinic for the 24- and 48-hour collections. Additional samples will be collected on Days 5 and 33.

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84, and 112. If a subject begins a steroid taper, additional photographs will be taken at the clinic visit during which the decision to begin the taper is made.

Subsequent visits will occur on Days 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42 and 56 for safety assessments, study drug dosing, sample collections, and other study procedures.

Subjects also will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

See Table 1 for a schedule of all study events. To assess safety and tolerability, subjects will undergo physical examinations (PEs; including weight), vital sign measurements, clinical (safety) laboratory tests, AE assessments, concomitant medication assessments, and electrocardiograms (ECG).

**Note**: No vaccinations may be given from within 2 weeks of screening through Day 56. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator.

# 4.4 Randomization and Blinding

This is an open-label study.

#### 5 STUDY POPULATION

#### 5.1 Target Population

This study will be conducted in approximately 16 male and female subjects (2 cohorts of 8 subjects each) with a confirmed diagnosis of pemphigus (vulgaris or foliaceus); however, a third cohort of up to 8 subjects may be added. Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled visits. The maximum number of subjects who may be enrolled in this study is 27 (24 + up to 3 replacements, as necessary). Within each dosing cohort, no more than 3 subjects may be enrolled with pemphigus foliaceus.

#### 5.2 Inclusion Criteria

A subject must meet the following criteria to be eligible for the study:

- 1. Willing and able to read, understand and sign an informed consent form;
- 2. Male or female  $\geq$  18 years of age;
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/ or skin lesions);
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal;
  - c. History of at least one positive tissue based test (biopsy, DIF)
- 4. Active disease: Lesions lasting > 2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion > 1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 antibodies, last dose > 12 months prior to screening;
  - b. If being treated with other immunosuppressants (i.e., azathioprine, mycophenolate mofetil or cyclosporine), must be on stable dose (< 10% change in dose) for 6 weeks prior to screening;
  - c. If being treated with corticosteroids, must be  $\leq 1 \text{mg/kg/day}$  of prednisone or equivalent and stable (< 10% change in dose) for 2 weeks prior to screening;

- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth
- 5. Body mass index (BMI)  $18.5 39.9 \text{ kg/m}^2$ ;
- 6. Has a negative pregnancy test (for women of childbearing potential) documented prior to the first dose of study drug;
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the Screening Period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through the final study visit.

#### 5.3 Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

- 1. Unable or unwilling to comply with the protocol;
- 2. Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ);
- 3. Positive for HIV or hepatitis C antibody;
- 4. Positive for hepatitis B surface antigen;
- 5. Active infection or history of recurrent infections;
- 6. IVIG treatment within 60 days of screening;
- 7. Received any cytotoxic (other than azathioprine) or mAb therapy in the 3 months prior to screening;

- 8. Any exposure to an investigational drug or device within 30 days prior to screening;
- 9. Plasmapheresis or immunoadsorption within 60 days of screening
- 10. Cellular therapy, including CAR-T, at any time prior to screening
- 11. Use of any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine within 3 months of screening;
- 12. Serum total IgG < 600 mg/dL;
- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (e.g., a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results);
- 14. Any vaccination within 2 weeks of screening

#### 6 STUDY PROCEDURES

#### 6.1 Informed Consent

All subjects must take part in the informed consent process. Adequate time must be allowed for the subject to ask questions and make a voluntary decision. No protocol-specific procedures, including screening procedures, are to be performed until the subject has signed and dated an IRB-approved ICF. Subjects may withdraw consent at any time. Participation in the study may be terminated at any time without the subject's consent as determined by the Investigator.

# 6.2 Demographics and Medical History

Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and eCRF. Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery and concomitant treatments, including relevant clinical response to past disease specific treatments and duration as well as dosing of such treatments.

### 6.3 Physical Examination

A complete physical examination will be performed as outlined in Table 1. The complete PE will include measurements of weight (in kg) and height (in cm; height to be measured only at screening visit) and a review of the following body systems:

- General appearance
- Head, eyes, ears, nose, and throat
- Neck
- Respiratory
- Cardiovascular
- Abdomen
- Neurologic
- Extremities
- Dermatologic
- Lymphatic

Any abnormal and clinically significant findings from the PE must be recorded in the appropriate eCRF. Findings at screening and Day 0 (pre-dose) will be recorded as medical history.

### 6.4 Pemphigus Disease Area Index (PDAI) Scoring

Pemphigus severity and disease activity will be measured using the PDAI. See Appendix B.

#### 6.5 Vital Sign Measurements

Vital sign measurements will be collected after the subject has been sitting for 5 minutes. Vital sign assessments will include measurements of sitting blood pressure (mm Hg), heart rate (beats per minute), respiration rate (breaths per minute), oral temperature (Celsius). Abnormal results are to be repeated after 5 minutes of rest. Pulse oximetry (%) also is to be measured. See Table 2 for timing window allowances with respect to measurement collection.

On Days 0, 7, 14, 21, and 28, vital sign measurements are to be obtained immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion. Details on the management of mild to moderate and severe infusion reactions can be found in Figure 1 and Figure 2. Abnormalities in vital sign measurements will be graded in severity per the NCI CTCAE scale Version 4.03.

Subjects should be seated quietly for at least 5 minutes in a chair with their backs supported, their feet flat on floor (legs uncrossed), and their arms bared on a hard surface, with the arm slightly abducted and bent, with palm up and the midpoint of upper arm at heart level. Correct cuff and bladder size should be utilized and the same cuff and arm should be used per subject throughout study.

#### 6.6 12-Lead Electrocardiogram (ECG)

Digital 12-lead ECG measurements will be obtained at screening, on Days 0 and 28 at 5 minutes after the completion of the infusion and at the Day 56 visit. Subjects who conduct their Day 12 visit at the investigative site, as opposed to an at-home nurse visit, will have an additional ECG performed. ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each 1 to 2 minutes apart. See Table 2 for timing window allowances with respect to performing ECG.

The following ECG parameters will be collected: PR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant.

Normal QTcF is  $\leq 450$  msec.

Abnormalities in the ECG that appear following therapy or that result in clinical signs and symptoms are considered clinically significant for the purposes of this study and will be recorded on the AE eCRF.

#### **6.7 Clinical Laboratory Measurements**

Collection time for all safety, PD, and exploratory labs are outlined in Table 1.

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and anti-drug antibody samples) will be performed using established methods by a central laboratory. Safety laboratory panels are defined as listed in Table 3. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and anti-drug antibody samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Full clinical safety lab draws will be collected at Screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 112. The total blood draw for each subject who completes the study at Day 112, will be approximately 433 mL. Please refer to the Laboratory Manual for more information.

Table 3: **Clinical Laboratory Panels** 

Syntimmune, Inc.

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| <ul> <li>CBC with differential and blood<br/>smear</li> <li>Erythrocyte Sedimentation Rate<br/>(ESR)</li> </ul> | <ul> <li>Albumin</li> <li>Alkaline phosphatase</li> <li>ALT</li> <li>AST</li> <li>BUN</li> <li>Calcium</li> <li>Carbon dioxide</li> <li>Chloride</li> <li>Creatinine</li> <li>Glucose</li> <li>LDH</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total and direct bilirubin</li> <li>Total protein</li> <li>Uric acid</li> <li>C-Reactive Protein</li> </ul> | <ul> <li>Appearance</li> <li>Color</li> <li>pH</li> <li>Specific gravity</li> <li>Ketones</li> <li>Protein</li> <li>Glucose</li> <li>Nitrite</li> <li>Urobilinogen</li> <li>Blood/hemoglobin</li> <li>Leukocyte esterase</li> <li>Bilirubin</li> <li>Microscopic examination of sediment: only if the results of the urinalysis dipstick evaluation are positive for blood/hemoglobin</li> </ul> |

#### Virology

- Hepatitis C
- Hepatitis B
- HIV
- VZV
- Tetanus

ALT = alanine aminotransferase; AST = aspartate aminotransferase; CBC = complete blood count; BUN = blood urea nitrogen; HIV = human immunodeficiency virus; LDH = lactate dehydrogenase; VZV = varicella-zoster virus

Abnormalities in clinical laboratory tests that are considered clinically significant are to be recorded on the AE electronic case report form (eCRF) page. Laboratory results will be graded using the NCI CTCAE, Version 4.03. If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as an SAE (see Section 11.3.1).

#### 6.7.1 Pregnancy Testing

Pregnancy testing will be performed for women of childbearing potential at screening and prior to first dose of SYNT001 on Day 0 and Days 56 and 112 (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing.)

# 6.7.2 Virology

Testing for HCV antibody, hepatitis B surface antigen, and HIV antibody will be performed at screening.

# 6.7.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

Samples for serum tetanus antibody and varicella-zoster virus antibody testing are to be collected at baseline (pre-dose, Day 0) and on Day 56 (Follow-Up visit). Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. Specifically, if the baseline VZV titer is above the detectable level, but tetanus is not, only the VZV antibody titer will be tested on Day 56. If the Day 56 results are below the baseline value, defined as greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 84; if still below the baseline value (or level of detection), the subject will be re-tested at Day 112. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112, will be referred to their primary care physician for further management.

### 6.7.4 Pharmacokinetics (PK) Sampling

Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. The actual time and date of each blood draw is to be recorded.

Study drug concentration will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-24}$ , and  $AUC_{0-\infty}$ .

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual

#### 6.7.5 Pharmacodynamic Sampling

PD samples will be collected for analyses throughout the study. On Days 0, 7, 14, 21, and 28, samples should be collected prior to infusion of study drug. Measurements for albumin PD biomarkers will be derived from the clinical safety laboratory results. Samples for each type of PD will be collected according to the schedule shown in Table 4.

Table 4: Pharmacodynamic/ Activity Assessments

| Parameter | Collection Timepoints |
|---|---|
| IgG, IgG subtypes (IgG1-4), IgA, IgM | Screening, and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, 56, 84 and 112. |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84 and 112 |
| Albumin | Screening, and Days 0, 7, 14, 21, 28, 33, 42, 56, 84 and 112 |
| Anti-Dsg (1 and 3) antibody titer | Screening, Days 0, 7, 14, 33, 56, 84 and 112 |
| <ul> <li>Complement component 3 (C3)</li> <li>Anti-epithelial cell antibody (AECA) levels by indirect immunofluorescence</li> </ul> | Days 0, 14, 33, 56, 84 and 112 |
| Exploratory biomarker (RNAseq, Urine IgG) | Days 0, 14, 33, 56, 84 and 112 |
| Immune phenotyping by flow cytometry for<br>measurement of CD3 <sup>+</sup> CD4 <sup>+</sup> T, CD3 <sup>+</sup> CD8 <sup>+</sup> T,<br>monocytes, NK cells and B cells | Days 0, 28 and 56 |
| Exploratory biomarker (FCGR2A SNP, via<br>buccal swab) | Day 0 |
| Exploratory pemphigus immune response<br>biomarkers | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84 and 112 |

See Table 2 for timing window allowances with respect to measurement collection. Detailed instructions for sample collection (including collection tubes) and preparation will be provided in a separate laboratory manual.

### 6.7.6 Immunogenicity Testing

Serum samples will be collected for immunogenicity analyses on Days 0 (pre-dose), 14, 28, 56, 84 and 112.

SYNT001 is being developed for the acute and chronic therapy of autoimmune disorders. Although SYNT001 is a humanized IgG4 monoclonal antibody, exposure to SYNT001 in clinical trials could result in the development of anti-drug antibodies (ADAs), with potential consequences ranging from neutralization or lessening of drug efficacy to safety consequences such as allergic reactions. Testing will first detect binding ADAs, then, for all confirmed positive samples, there will be testing for neutralizing effects.

Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

### 6.8 Study Drug Administration

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute IV infusions of SYNT001 10 mg/kg or up to 30 mg/kg. SYNT001 will be given as a 250-mL IV infusion over 1 hour using a 0.2-micron, inline filter. Based on review of safety data, as well as available and relevant PD results, and clinical outcomes of Cohort 1, a decision about proceeding with Cohort 2 will be made. Based on review of all safety data, available PD results, and clinical outcomes of these 2 cohorts, a third cohort of 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

| Cohort No. | Study Drug | Dose Level<br>(mg/kg/dose) |
|------------|------------|----------------------------|
| 1 | SYNT001 | 10 mg/kg |
| 2 | SYNT001 | 30 mg/kg |

See Section 9.1 for dosing schedule.

#### 6.9 Prior and Concomitant Medications

All medications a subject receives within 14 days prior to enrollment through the end of the study will be documented on the source document and eCRF. A history of treatments taken for primary disease, even if not taken within the 14 days prior to enrollment, will be collected.

Note: No vaccinations may be given from within 2 weeks of screening through Day 56. Following Day 56, subjects may receive vaccinations at the discretion of the Investigator.

#### 6.10 Adverse Event Assessments

Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form and continuing through the last study visit. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE.

Clinical AEs will be graded using the NCI CTCAE, Version 4.03 (Appendix A).

**Note**: AEs resulting in a subject's permanent discontinuation from the study, regardless of seriousness or relationship to study drug, MUST be promptly reported to the sponsor. Additionally, subjects must be followed until return to normal and/or resolution of the AE.

See Section 11 for more information.

### 6.11 Photographs

On Day 0 photographs will be taken of active lesions. Follow-up photographs will be taken of the same areas on Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

### 6.12 Skin Biopsy

Optional skin biopsy samples from lesional or non-lesional skin will be collected on Day 0 predose and on Days 1, 2, 14, 33, 56 and 84 to analyze SYNT001 levels.

#### 7 STUDY ASSESSMENTS

#### 7.1 Screening Period: Day -14 to Day -1

Informed consent must be obtained before any study-specific samples are taken or study-specific tests or evaluations are conducted. The following assessments at the screening visit are to occur within 14 days before dosing. Study eligibility will be based on satisfying all the study inclusion and exclusion criteria.

At the screening visit, information will be collected and subjects will have clinical evaluations as follows:

- Informed consent (Section 6.1)
- Medical history and demographic data (Section 6.2)
- Review inclusion and exclusion criteria (Section 5.2, Section 5.3)
- Complete PE, including height and weight (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Section 6.6)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section
- Pregnancy test (Section 6.7)
- Hepatitis and HIV screen (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.2 **Enrollment and First Treatment: Day 0**

Study Day 0 is defined as the date the subject is administered their first dose of study drug. On Day 0, subjects will be asked to come to the clinic and the following procedures will be performed prior to the first dose of study drug:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)

- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody (Section 6.7)
- PDAI Score (Section 6.4)
- PK baseline sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - FCGR2A SNP, via buccal swab
  - RNAseq
  - Urine IgG
  - Immune phenotyping
  - Exploratory pemphigus immune response biomarkers
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.3 Follow-up: Day 1

On Day 1 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.4 Follow-up: Day 2

On Day 2 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.5 Follow-up: Day 5

On Day 5 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 0), subjects may return to the clinic or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.6 Treatment Day 7 (Dose 2)

On Day 7 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral

- temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.7 Dose 2 Follow-up Day 12

On Day 12 ( $\pm$  6 hours) the subject may return to the clinic, or be visited by at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- If visit performed at the study site: 12-Lead ECG to be obtained in triplicate (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.8 Treatment Day 14 (Dose 3)

On Day 14 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)

- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg (1 and 3) antibody titer
  - CIC
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Optional skin biopsy (Section 6.12)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)

AE assessment (Section 6.10)

### 7.9 Dose 3 Follow-up Day 19

On Day 19 ( $\pm$  6 hours) the subject may return to the clinic, or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.10 Treatment Day 21 (Dose 4)

On Day 21, ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- PDAI Score (Section 6.4)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion

Protocol SYNT001-103

and at completion of the infusion (Section 6.5)

- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.11 Treatment Day 28 (Dose 5)

On Day 28 ( $\pm$  6 hours), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam (Section 6.3)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature); to be measured immediately prior to the infusion (Section 6.5)
- Pulse oximetry (to be measured immediately prior to the infusion) (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (collected just prior to the start of the study drug infusion; record collection date and time for each PK sample) (Section 6.7)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion) (Section 6.7)
- PD sample collection (collected just prior to the start of the study drug infusion) (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Immune phenotyping
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug) (Section 9)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Pulse oximetry will be measured at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion (Section 6.5)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature): 30 minutes, 1 hour and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Pulse oximetry: 30 minutes, 1 hour and 2 hours following completion of the infusion (Section 6.5)
- PK sample collection at 5 minutes and 2, 4, 6 hours after the end-of-study drug infusion; record collection date and time for each PK sample (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion (Section 6.6)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.12 Follow-up Day 29

On Day 29 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

# 7.13 Follow-up Day 30

On Day 30 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- PK sampling (record collection date and time) (Section 6.7)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.14 Follow-up Day 33

On Day 33 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 28), subjects will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PK sampling (record collection date and time) (Section 6.7)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

### 7.15 Follow-up Day 42

On Day 42 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.16 Follow-up Day 56

On Day 56 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- 12-Lead ECG (to be obtained in triplicate after 5 minutes of rest in the sitting position) (Section 6.6)
- Serum tetanus antibody and VZV antibody; Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC

- Anti-Dsg (1 and 3) antibody titer
- C3
- AECA
- RNAseq
- Urine IgG
- Immune phenotyping
- Exploratory pemphigus immune response biomarkers
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 7.17 Follow-up Day 84

On Day 84 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Serum tetanus antibody and VZV antibody testing if required. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Optional skin biopsy (Section 6.12)
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

## 7.18 Follow-up Day 112 (End-of-Study) or Early Termination Visit

On Day 112 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam (Section 6.3)
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest (Section 6.5)
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis) (Section 6.7)
- Pregnancy test (Section 6.7)
- Serum tetanus antibody and VZV antibody testing if required. See Section 6.7.3 for additional information.
- Immunogenicity sample collection (Section 6.7)
- PDAI Score (Section 6.4)
- PD sample collection (Section 6.7)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titer
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Photography (Section 6.11)
- Concomitant medication assessment (Section 6.9)
- AE assessment (Section 6.10)

#### 8 REMOVING SUBJECTS FROM STUDY

Every reasonable effort will be made to keep the subject in the study; however, if a subject is withdrawn from the study, every effort will be made by the Investigator to complete and report the reasons for withdrawal as thoroughly as possible. The reason(s) for termination must be clearly documented on the appropriate page of the eCRF. Once a subject discontinues from the study for any reason, every effort will be made to collect all clinical and laboratory data as scheduled for the Early Termination Visit (See Table 1). A termination eCRF must be completed for all enrolled subjects.

### 8.1 Subject Withdrawal

A subject's participation in the study may be prematurely discontinued for any of the following reasons:

- 1. The subject wishes to withdraw from the study.
- 2. Request by a regulatory agency (e.g., Institutional Review Board).
- 3. Subject experiences a significant or intolerable AE.
- 4. The subject experiences a significant adverse change in vital signs, PE findings, or a clinical laboratory parameter.
- 5. The subject has a need for a concomitant medication that is not permitted by the study protocol.
- 6. The subject experiences generalized impairment or mental incompetence that would result in the subject being unable to understand his or her participation in the study.
- 7. If, in the Investigator's medical judgment, further participation would be injurious to the health and well-being of the subject, or is not in the best interest of the subject.
- 8. Administrative reasons, such as subject non-compliance or a major protocol violation.

Subjects who are withdrawn from this study due to an AE determined to be related to study drug are to be followed until there is either:

- Resolution or stabilization of the AE determined to be related
- The subject is lost to follow-up
- The event is otherwise explained

If there is a persistent AE contributing to discontinuation that is determined to be related to SYNT001, subjects must be followed with appropriate medical management until resolution or stabilization.

A reasonable effort should be made to contact any subject lost to follow-up during the study to complete assessments and retrieve any outstanding data. If the subjects are unreachable by telephone after three (3) attempts, the minimum of a registered letter should be sent requesting that contact be made with the Investigator to report survival information.

## 8.2 Study Discontinuation

Syntimmune Inc. has the right to terminate or to stop the study at any time. Reasons for study discontinuation may include, but are not limited to the following:

- The incidence or severity of AEs in this or other related studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Drug supply issues
- Excessive subject self-withdrawal
- Significant protocol violations (e.g., violation of eligibility criteria, dosing errors, missing data for study endpoint analysis)

### 8.3 Replacements

Enrolled subjects withdrawn for a reason other than an AE will be replaced if they have not been dosed or have only received one dose of study drug at the time of discontinuation, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled study visits.

# 8.4 Stopping Rule

### 8.4.1 Dose-Escalation Stopping Rule

Dose escalation decisions will be made by a Dose Escalation Committee (DEC) and will be based on safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities, AEs, SAEs, and total IgG levels.

Dose-limiting toxicity (DLT) will be defined generally as severe (Grade 3) AEs occurring in  $\geq$ 2 subjects that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort (8 total subjects per cohort) have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. If the dose-escalation stopping rule is met during Cohort 1 (10 mg/kg) all safety data and all available pharmacodynamics will be reviewed and the cohort may resume (if applicable) or a new cohort may be added at a dose at least 50% lower than the 10 mg/kg dose. If the stopping rule is not met in Cohort 1, dose-escalation may proceed up to a maximum of 30 mg/kg. If the dose-escalation stopping rule is met for the first time during Cohort 2, all safety data and all available pharmacodynamics will be reviewed and the cohort may resume (if applicable) or a new cohort may be added at a dose a minimum of 30% lower than the Cohort 2 dose. If the stopping rule is not met in Cohort 2, dose-escalation may proceed up to a maximum of 45 mg/kg; however, this cohort may also receive a dose equal to or less than 30 mg/kg based on evaluation of all safety and pharmacodynamic data.

### 8.4.2 Study Stopping Rule

If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects.

#### 8.4.3 Individual Stopping Rule

Dosing for any individual subject will be discontinued (i.e., no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related non-SAE adverse event that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) suggest that it could be unsafe to administer further study drug to that subject. Additionally, a subject will be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus.

#### 9 STUDY DRUG

For detailed information regarding SYNT001 preparation and administration, refer to the Pharmacy Manual.

#### 9.1 SYNT001

SYNT001 is provided in vials containing 5 mL SYNT001 (extractable volume) at a nominal concentration of 50 mg/mL. The product is supplied as a liquid at pH  $6.5 \pm 0.5$ . SYNT001 is diluted in Dextrose 5% in Water (D5W) to prepare the solution for infusion. SYNT001 will be infused via IV in 250 mL over 1 hour using a 0.2-micron, inline filter.

Two cohorts of 8 eligible subjects each will receive 5 once-weekly 60-minute infusions of SYNT001 in planned doses of 10 mg/kg or 30 mg/kg. Based on review of safety, PD, and clinical outcomes of these two cohorts, a third cohort of up to 8 subjects may be treated at another dose, with a maximum dose of 45 mg/kg, but may also be lower than 10 mg/kg or between 10 and 30 mg/kg, inclusive.

The specification for host cell DNA in SYNT001 is < 2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing is limited to 5000 mg of SYNT001. Therefore, the maximum subject weight allowed for enrollment into the 30 mg/kg dose cohort is 166 kg and the maximum subject weight allowed for enrollment into the highest dose possible in this study (45 mg/kg)is 111 kg.

### 9.2 Cohort Dosing

Cohorts will be dosed sequentially beginning with Cohort 1. The first 2 subjects will be dosed at least 24 hours apart. A review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject. A review of the 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining 6 subjects in the cohort. Cohort 2, and Cohort 3 if added, will be dosed per the same schedule

#### 9.3 Timing of Dosing

On Days 0, 7, 14, 21, and 28, subjects will receive a 60-minute IV infusion of SYNT001 in the morning. The date and time the dose is administered will be recorded.

### 9.4 Identity of Investigational Products

All supplies of SYNT001 will be supplied by Syntimmune and must be stored refrigerated (2°C to 8°C/36°F to 46°F) in the carton and protected from light, in a securely locked area, accessible

to authorized persons only, until needed for dose preparation. Qualified site personnel will inventory the investigational product received and will maintain records of disposition of the drug, including dates, quantity and use.

### 9.5 Investigational Product Retention at Study Site

The Investigator (or designee) is responsible for maintaining accurate accountability records of the investigational product throughout the clinical study. All study drug received at the site must be inventoried and accounted for in an accountability log provided by the Sponsor. All dispensing and accountability records will be available for Sponsor review. Study drug accountability will be verified during on-site monitoring visits.

Upon the completion or termination of the study, and upon written authorization from the Sponsor, or its representative, all unused and/or partially used study drug should be returned or destroyed at the investigational site, as specified by Sponsor. It is the Investigator's responsibility to ensure that the Sponsor, or its representative, has provided written authorization that procedures for proper disposal of the study drug have been established, and that appropriate records of the disposal are documented and maintained. No unused study drug may be disposed until fully accounted for by the Sponsor monitor (or designee)

## 9.6 Warnings and Precautions

**Note:** Subjects must not receive any vaccinations from within 2 weeks of screening until Day 56.

#### 9.6.1 Infusion Reaction

SYNT001 will be given as an IV infusion over 1 hour. As with all mAbs administered by IV infusion, infusion reactions are possible. In nonclinical testing of SYNT001 in NHPs, clinical observations were limited to infusion reactions due to the immunogenicity of SYNT001 in NHPs. These reactions included transient emesis/vomitus which typically occurred within 1 hour of dosing at all dose groups, but only after the third weekly infusion following the development of ADAs. Transient histamine-type responses were noted 30 minutes post-dose in some animals in all dose groups, but only following the third weekly infusion as above. These reactions were consistent with a histamine reaction (decreased activity, periocular swelling, erythema, facial flushing, eyelids partially/completely closed, and/or generalized weakness). With the exception of vomitus/emesis and red skin discoloration associated with injection or blood draw sites, these observations spontaneously resolved within 1-hour post-dose. Subsequent pretreatment with intramuscular diphenhydramine prevented further histamine-type reactions. All doses of SYNT001 were administered by bolus infusion over approximately 5 minutes in the NHP

studies. However, all of the observed infusion reactions (including vomitus/emesis and histamine-type reactions) associated with ADAs are not at all predictive of what may occur in humans (Bugelski and Treacy, 2004; Ponce et al., 2009) and furthermore, are not considered relevant to predicting responses in humans [ICH S6(R1) 2011].

Typically, infusion reactions to monoclonal antibodies observed in human studies develop within 30 minutes to 2 hours after the initiation of drug infusion, although symptoms may be delayed for up to 24 hours. Most are mild in severity, although severe and even fatal reactions can occur.

### Guidelines for Grading and Management of Allergic or Infusion-Related Reactions

Allergic and/or infusion-related reactions include hypersensitivity reactions and cytokine release syndromes. These reactions are experienced by patients during or within hours of the infusion of monoclonal antibody therapy. Symptoms can include flushing, alterations in heart rate and blood pressure, dyspnea, bronchospasm, back pain, fever, urticaria, edema, nausea, and all types of rashes. Anaphylaxis is recognized as a severe, life-threatening, generalized, or systemic reaction. This is a medical emergency characterized by rapidly developing life-threatening airway and/or breathing and/or circulation problems usually associated with skin or mucosal changes.

Management of Grade 1 infusion reactions include interrupting the infusion or decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen, either alone or in combination, depending on the subject's signs and symptoms. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 administration.

Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. See Figure 1 and Figure 2 for details on the management of Grade 2 and Grade 3 or higher infusion reactions. The severity of and management of allergic or infusion-related reactions will be graded and managed using NCI CTCAE Version 4.03 (see Table 5).

Figure 1: Management of Moderate (Grade 2) Infusion Reactions



If symptoms and signs resolve completely either spontaneously or after administration of diphenhydramine with or without hydrocortisone, consider rechallenge:

Wait at least 20 minutes following medication administration before commencing rechallenge at an infusion rate of 50% or less of the initial infusion rate or

Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 administration.

Syntimmune, Inc.


Amendment 3.0 Final 10 October 2017

Figure 2: Management of Severe (Grade 3 or higher) Infusion Reactions

Subject presents with any of the below:

- Urticaria
- Airway threatened by angioedema
- Angioedema: Lip, mouth, facial swelling
- Respiratory compromise wheezing, dyspnea, stridor or hypoxia (O2 saturation < 90%)
- BP < 90 mmHg SBP or >30% decrease from patient baseline



Start basic life support:

- High oxygen flow
- On bed, head down, legs up
- Large bore IV cannula, 1 L normal saline STAT
- Initiate vital signs at least every 15 minutes



Consider (under medial direction):

Epinephrine 1:1000

• 0.3 mg (0.3 mL) IM into lateral thigh



Airway Threatened: Nebulized epinephrine 1:1000, 3–5 mL (3–5 mg)

**Bronchospasm:** Nebulized salbutamol 5 mg

(Wheeze or Hypoxia) Consider: Intubation / nebulized epinephrine

**Hypotension:** Place on cardiac monitor

(Systolic BP <100 mmHg) Further epinephrine 1:1000, 0.3 mg IM and

IV normal saline bolus 20 mL/kg STAT as needed

Have vasopressin on hand



Transfer to Emergency Room/ICU Observe until all symptoms resolved.
Table 5: Grading and Management of Allergic or Infusion-Related Reactions

| Adverse<br>Event | Grade | | | | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| Infusion-<br>Related<br>Reaction | Mild transient<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Allergic<br>Reaction | Transient<br>flushing or<br>rash, drug<br>fever<br>< 38.0°C.<br>Intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Anaphylaxis | - | - | Symptomatic<br>bronchospasm, with or<br>without urticarial;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Cytokine<br>release<br>syndrome | Mild<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤ 24 hours | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>pressor or<br>ventilator<br>support<br>indicated | Death |

Abstracted from NCI CTCAE Version 4.03.

#### 9.6.2 Potential Immune Effects

An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels after a single dose and further decreases after multiple doses up to a 70% to 80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within 30% of baseline levels observed at pretreatment occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.

Given the normal adult range of IgG of 500 to 1600 mg/dL (Agarwal and Cunningham-Rundles, 2007; Furst, 2009; Gonzalez-Quintela et al., 2008; Jolliff et al., 1982; Keystone et al., 2007; McMillan et al., 1997; van Vollenhoven et al., 2013), with a mean of 1150 mg/dL, a 50% decrease in the mean would be to 575 mg/dL and a 50% decrease from the low end of the normal range used for the inclusion criteria of 600 mg/dL would be to 300 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 120 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency (Ameratunga et al., 2013), the levels will be transient. Further, as reported for other therapies used for pemphigus, the temporary (ie, less than 4 months) depletion of IgG (up to 95% reduction of total IgG as seen with immunoadsorption) does not appear to impart an increased risk of infection (Eming and Hertl, 2006; Furst, 2009; Keystone et al., 2007; Schmaldienst et al., 2001; van Vollenhoven et al., 2013). Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to reverse the low IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

An antibody blocking FcRn is expected to also down modulate innate and adaptive immunity and the catabolism of IgG-containing immune complexes (IC). Specifically, it is expected that anti-FcRn will promote the clearance of IgG-containing ICs and the effects of these IC on stimulating innate immune cell production of inflammatory cytokines (e.g., IL-12, interferon-γ, and tumor necrosis factor [TNF]) and inhibit the processing and presentation of antigens contained within IC and thus the antigen-specific activation of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells. Therefore, subjects with pre-existing conditions that are dependent upon IgG antibodies, such as chronic infections (e.g., HIV, HBV or HCV), will be excluded from this study, as will subjects with active infection in general.

SYNT001 administration could decrease the level of protective antibodies from prior vaccinations. Protective antibody levels for tetanus and varicella-zoster virus (chickenpox) are to be tested in accordance with Section 6.7.3.

#### 10 CONCOMITANT MEDICATION AND TREATMENT

All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. Premedication is discouraged as prophylaxis against AEs or infusion reactions unless medically indicated from either past medical history, prior infusion reactions or AEs resulting from SYNT001 infusions.

Use of the following treatments will not be permitted during the study unless otherwise specified:

- Rituximab or other anti-CD20 antibody
- Monoclonal antibodies other than study drug
- Any immunosuppressive drugs apart from corticosteroids, azathioprine, mycophenolate mofetil, or cyclosporine.
- Topical steroids
- Any dietary herbal supplements
- Any investigational drug or device
- Any vaccinations through Day 56. Following Day 56, subjects may be vaccinated at the discretion of the Investigator.

If over a period of at least two weeks on study drug, a subject on corticosteroids shows the absence of new lesions and significant healing of lesions that existed at study baseline, a slow corticosteroid taper may be started as per the following suggested schedule

- If on > 30 mg of prednisone per day, decrease by 10 mg every two weeks until a dose of 30 mg per day then decrease by 5 mg every two weeks
- If on < 30 mg of prednisone per day, decrease by 5 mg every two weeks

In cases in which concomitant medications are used, details to be recorded include the following: medication name, start date and time, stop date and time, dose, route, frequency, and reason for use. The concomitant medication names are to be coded using the World Health Organization (WHO) Drug Dictionary (WHO-DD March 2013, Type B2 or later) and classified by anatomical therapeutic chemical (ATC) categories.

#### 11 SAFETY

# 11.1 Safety Parameters

Clinical and laboratory AEs will be graded using the NCI CTCAE; Version 4.03 (See Appendix A).

Subjects will be monitored throughout the treatment and follow-up period for occurrence of AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status, vital sign measurements, and laboratory data (including PD). Safety parameters to be measured/assessed include PEs, vital sign measurements, hematology, serum chemistries, urinalysis, and ECG.

#### 11.2 Adverse Event Definition

An AE is defined as any untoward medical occurrence in a clinical trial subject associated with the use of a drug, whether considered drug related. An AE can be an unfavorable and unintended sign (e.g., an abnormal laboratory value finding), a symptom, or a disease temporally associated with the use of a drug, without judgment as to causality. An AE can arise from use of the drug (e.g., use in combination with another drug) and from any route of administration, formulation or dose, including an overdose. An AE also includes, but is not limited to, any clinically significant worsening of a pre-existing condition. Examples include:

- Any sign, symptom, physical finding, or laboratory result that has worsened in nature, severity or frequency compared to baseline;
- Reactions from an investigational drug, including those occurring because of an overdose, abuse of the study drug, withdrawal phenomena, sensitivity or toxicity;
- Concurrent illness that was not present or worsens in nature, severity, or frequency compared to baseline;
- Injury or accident; and/or
- Exacerbation of a pre-existing condition.

For data collection, all untoward events that occur after informed consent through the last study visit are to be recorded on eCRFs by the investigational site.

While pregnancy alone is not considered as an AE or SAE, any pregnancy complication(s) should be recorded as an AE(s) or SAE(s) (if applicable). Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions (see below). Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. If a female subject becomes pregnant during the conduct of the study, the Investigator must notify the Sponsor according to the procedures provided in Section 11.3.8).

# 11.3 Evaluating Adverse Events

The Investigator will determine the seriousness, intensity, and causality of an AE associated with the use of the study drug (i.e., events where there is a reasonable possibility that the event may have been caused by the study drug) based on the definitions that follow.

#### 11.3.1 Serious Adverse Events

(Notify Medpace Safety within 24 hours; document on eCRF)

The SAE definition and reporting requirements are in accordance with Title 21 Part Code of Federal Regulations (CFR) 312.32 and the Guidance for Industry and Investigators Safety Reporting Requirements for Investigational New Drug (INDs) and Bioavailability /Bioequivalence Studies.

SAE: An AE is considered "serious" if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:

• <u>Death:</u> This includes any death that occurs while the subject is "on study" through the last study visit.

**Note**: Death is an outcome of an AE, and not an AE. The event(s) that caused death (e.g., illness, accident) is the SAE. Death due to any other cause(s) must also be reported as an outcome of the reportable SAE.

- <u>Life-threatening adverse drug event:</u> An AE or suspected adverse reaction is considered "life threatening" if, in the view of either the Investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.
- Inpatient hospitalization or prolongation of existing hospitalization:

In the absence of an AE, the Investigator should not report hospitalization or prolongation of hospitalization. This is the case in the following situations:

- Hospitalization or prolongation of hospitalization is needed for a procedure required by the protocol
- Hospitalization or prolongation of hospitalization is part of routine procedure followed by study center

- Hospitalization for survey visits or annual physicals
- Hospitalization for observation with release within 24 hours

In addition, a hospitalization planned before the start of the study for a pre-existing condition, which has not worsened, does not count as an SAE.

- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Congenital anomaly/birth defect
- <u>Important medical event:</u> An event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 11.3.2 Overdose

An overdose is defined as a significant variation from the recommended/scheduled dosage for a product. The dosing for this study will be conducted in a controlled clinical setting and an overdose is not anticipated. However, in the event of an accident, for this study, an overdose of SYNT001 is considered a dose that is two-fold higher than the intended dose for the subject.

#### 11.3.3 Non-Serious Adverse Events

(Document on eCRF)

All other AEs, not fulfilling the previous definitions, are classified as non-serious.

#### 11.3.4 Protocol-Related Adverse Events

AEs that are not test drug related may nevertheless be considered by the Investigator or the Medical Monitor to be related to the conduct of the clinical study. That is, the event may be related to the fact that a subject is participating in the study. For example, a protocol-related AE may be an event that occurs during a screening period or that is related to a procedure required by the protocol.

#### 11.3.5 Assessment of Causality

A medically qualified Investigator must assess the relationship of any AE (including SAEs) to the use of the investigational product, as related or not related, based on clinical judgment and using all available information, and may include consideration of the following factors:

- Possible alternative causes of the AE, including the disease under treatment, pre-existing conditions, concomitant use of other drugs, and presence of environmental or genetic
- The temporal association between drug exposure and onset of the AE.
- Whether the manifestations of the AE are consistent with known actions or toxicity of the investigational product.
- The AE resolved or improved with decreasing the dose or stopping use of the investigational product (dechallenge). Judgment should be used if multiple products are discontinued at the same time.

The causal relationship between the study medication and the AE will be assessed using one of the following categories:

**Not Related:** Factors consistent with an assessment of Not Related include:

- Temporal relationship is lacking (e.g., the event did not occur within a reasonable time frame following administration of the study medication); or
- Other causative factors more likely explain the event (e.g., a pre-existing condition, other concomitant treatments).

**Related:** Factors consistent with an assessment of Related include:

- There is a positive temporal relationship (e.g., the event occurred within a reasonable time frame following administration of study medication); or
- The AE is more likely explained by the investigational product than by another cause (i.e., the AE shows a pattern consistent with previous knowledge of the investigational product or the class of the investigational product)

#### 11.3.6 **Recording Adverse Events**

All AEs (including SAEs) are to be accurately recorded on the Adverse Event page of the subject's eCRF. The severity of each AE will be graded using the NCI CTCAE, Version 4.03. The date of onset as well as the end date of the event also should be recorded or the event should be entered as "ongoing". In addition, the method used to treat the AE and the outcome of the AE also will be noted. The Investigator will assess the relationship of the event to study drug.

#### 11.3.7 **Planned Hospitalization**

A hospitalization planned by the subject prior to the first dose of study medication is considered a therapeutic intervention and not the result of a new SAE and should be recorded as medical

history. If the planned hospitalization or procedure is executed as planned, the record in the subject's medical history is considered complete. However, if the event/condition worsens during the trial, it must be reported as an AE.

#### 11.3.8 Reporting Pregnancies

If a female subject or the female partner of a male subject becomes pregnant during the course of the study, the Investigator must report the pregnancy to the Medpace Safety using the **Pregnancy Reporting Form** within **24 hours** of becoming aware of the event. The Investigator must obtain consent to collect pregnancy information (including the status of the newborn, if applicable).

If some of the information required for completion of the Pregnancy Reporting Form is unavailable at the time of the initial report, follow-up reports will be completed and submitted within 24 hours of becoming aware of the new information. Any pregnancy will be followed through delivery for the observation of any SAEs. Any SAE that occurs during pregnancy must be recorded on the SAE report form in the EDC system (e.g., maternal serious complications, therapeutic or spontaneous abortion, ectopic pregnancy, stillbirth, neonatal death, congenital abnormality, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs (See Section 11.3.9).

#### 11.3.9 Serious Adverse Event Reporting

# 11.3.9.1 Governing Regulatory Requirements

Compliance with this request for prompt reporting is essential in that the sponsor is responsible for informing the US Food and Drug Administration (FDA) and other regulatory authorities as well as all other participating Investigators of the event.

Under FDA ruling (US Code of Federal Regulations, Title 21 CFR Part 312.32) and the ICH Guidelines for Clinical Safety Data Management Definitions and Standards for Expedited Reporting, the sponsor is required to submit written documentation, in the form of a safety report, detailing:

- Any event associated with the use of the drug, that is both serious and unexpected, or
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects, including reports of <u>mutagenicity</u>, <u>teratogenicity</u>, <u>or carcinogenicity</u>.

Written submission must be made by the sponsor to the FDA as soon as possible and in no event later than 15 calendar days after the sponsor's initial notification of the event. The sponsor shall also inform all Investigators.

# 11.3.9.2 Time Frame for Reporting

Any death, SAE or pregnancy experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, , must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee).

Contact information for **SAE** reporting:



Additionally, the Investigator will be able to contact the **Medical Monitor**:



#### 11.3.9.3 Information to be Provided by the Investigator

SAEs must be recorded on the SAE form in the EDC system. This requirement includes all SAEs that occur after informed consent through the last study visit.

The minimum information required for SAE reporting includes identity of Investigator, site number, subject number, an event description, SAE term(s), onset date, the reason why the event is serious (i.e., the seriousness criteria) and the Investigator's assessment of the relationship of the event to study treatment. Additional SAE information including medications or other therapeutic measures used to treat the event, action taken with the study treatment due to the event, and the outcome/resolution of the event will be recorded. Paper forms for reporting SAEs will be provided to the study sites as back-up in case the EDC system is not accessible.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. Furthermore, the Investigator may be required to provide supplementary information as requested by Syntimmune or designee.

When reporting an SAE, the following additional points should be noted:

When the diagnosis of an SAE is known or suspected, the Investigator should report the
diagnosis or syndrome as the primary SAE term, rather than as signs or symptoms. Signs
and symptoms may then be described in the event description. For example, dyspnea
should not be used as an SAE term if the diagnosis, which caused the dyspnea, is known
to be malignant pleural effusion.

- Death should not be reported as an SAE, but as an outcome of a specific SAE, unless the event preceding the death is unknown. In the exceptional case where the events leading to death are unknown, then death may be used as an event term. If an autopsy was performed, the autopsy report should be provided.
- While most hospitalizations necessitate reporting of an SAE, some hospitalizations do not require SAE reporting, as follows:
  - Elective or previously scheduled surgery, e.g., a previously scheduled ventral hernia repair
  - Procedures for pre-existing conditions that have not worsened after initiation of treatment
  - Pre-specified study hospitalizations for observation
  - Events that result in hospital stays of less than 24 hours and that do not require admission, e.g., an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics
- SAEs must, however, be reported for any surgical or procedural complication resulting in prolongation of the hospitalization.

#### 11.3.10 Regulatory Reporting

Syntimmune (or designee) will process and evaluate all SAEs as soon as the reports are received. For each SAE received, Syntimmune will decide as to whether the criteria for expedited reporting have been met.

Syntimmune (or designee) will submit SAEs that meet the criteria for expedited reporting to the regulatory authorities in accordance with local regulations governing safety reporting. Reporting of SAEs by the Investigator to his or her IRB will be done in accordance with the standard operating procedures and policies of the IRB. Adequate documentation must be maintained showing that the IRB was properly notified.

# 11.3.11 Follow-up Information on a Serious Adverse Event (SAE)

Appropriate diagnostic tests should be performed and therapeutic measures, if indicated, should be instituted. Appropriate consultation and follow-up evaluations should be carried out until the event has returned to baseline or is otherwise explained by the Investigator.

If all required information on the SAE form is not available at the time of the initial report, follow-up information will be completed in the EDC system.

# 11.4 Other Safety Considerations

# 11.4.1 Laboratory Data

All laboratory data obtained during the study should be reviewed. Any abnormal value that leads to a change in subject management (e.g., requirement for additional medication or monitoring) or is of clinical significance by the Investigator should be reported as an AE and/or SAE as appropriate, unless this value is consistent with values obtained before entry into the study.

#### 11.4.2 Medication Errors

Any medication error that results in an AE, even if it does not meet the definition of serious, requires reporting within 24 hours to the safety Medical Monitor.

#### 11.4.3 Follow-Up of Adverse Events

Any SAE or AE assessed as related to study drug must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. The Investigator will follow all drug related AEs until there is a return to the subject's baseline condition, or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary. The status of all AEs will be documented as of the last study visit.

Where a diagnosis is possible, it is preferable to report this diagnosis rather than a series of terms (signs/symptoms) relating to the diagnosis.

# 11.5 Safety Monitoring for Dose Escalation

Following dosing in each cohort, all safety/tolerability data (e.g., PEs, vital signs [including pulse oximetry], clinical safety laboratory tests, ECGs and AE/SAE assessments) as well as any available and relevant PD data collected through Day 42 will be reviewed by the DEC. A decision to escalate to the next cohort will be made. The recommendation may be to continue to

the next scheduled dose level, discontinue the study or to modify dosing to a dose less than the current dose or higher than the current dose but lower than the next planned dose.

#### 12 STATISTICAL CONSIDERATIONS

All descriptive and inferential statistical analyses will be performed using the most recently released and available Statistical Analysis System (SAS) software, unless otherwise noted. Missing data will not be imputed unless otherwise stated. All clinical data captured will be provided in data listings. A Statistical Analysis Plan (SAP) and a Pharmacokinetic Analysis Plan (PAP) will be finalized prior to database lock.

# 12.1 General Design

All data for enrolled subjects will be presented in data listings by subject number.

Continuous data will be described using descriptive statistics: number of observations (n), mean, standard deviation (SD), median, minimum, and maximum. Frequencies and percentages will be used for summarizing discrete (categorical) data. When categorical data are presented, the percent will be suppressed when the count is zero to draw attention to the non-zero counts. The denominator for all percentages, unless otherwise specified, will be the number of subjects in the specified analysis population.

#### 12.2 Sample Size Justification

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

#### 12.3 Statistical Considerations

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). The SAP may modify the plans outlined in the protocol; any deviations from the previously described statistical plan will be described and justified in an SAP amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate and will be described in the SAP. Methods of handling of missing data for different endpoints will be further specified in the SAP. In general, where individual data points are missing because of insufficient samples, dropouts, or other reasons, the data will be analyzed based on reduced denominators unless specified otherwise in the SAP.

Results will be summarized by cohorts.

# 12.3.1 Study Populations

Three populations will be employed in the analysis of study data:

• The **intent-to-treat (ITT)** population will consist of all subjects who have received at least one dose of study drug. All safety analyses will be performed on the ITT population.

- The **PK** population will consist of all subjects who receive at least one dose of study drug and have sufficient post-dose blood samples to obtain PK parameters.
- The **PD** population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.

Primary safety analyses will be performed on the ITT population. Demographics, subject disposition, and screening and baseline characteristics will be summarized for the ITT, PK, and PD populations, where appropriate.

#### 12.3.2 Subject Accountability, Demographics, and Baseline Characteristics

Subject disposition, demographic information and baseline characteristics will be presented. Any discrepancy between treatment to be given and treatment received will be accounted for in these displays.

#### 12.3.3 Concomitant Medications

Concomitant medications will be coded using WHO Drug Dictionary (WHO-DD March 2013, Type B2 or later) and the data will be summarized and presented in tables and listings.

# 12.4 Planned PK Analysis

Study drug concentrations will be used to calculate the following PK parameters:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ , and  $AUC_{0-24}$  and  $AUC_{0-\infty}$ . PK parameters will be determined using noncompartmental method(s). Descriptive statistics of PK parameters for SYNT001 will include mean, SD, coefficient of variation (CV), median, minimum, and maximum.  $T_{max}$  will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after  $log_{10}$  transformation of PK parameters.

For calculation of mean concentrations and generation of mean concentration-time profiles, all below the limit of quantification (BLQ) values will be set to zero except when an individual BLQ falls between 2 quantifiable values, in which case it will be omitted.

If there are values above the BLQ, but too sparse to allow full analysis, descriptive statistics will be performed on available values.

# 12.5 Safety Data

Safety observations and measurements include AEs, safety laboratory tests, vital sign measurements, PEs, and ECGs.

Treatment-emergent AEs will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least 1 occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

AEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject, cohort, and overall per SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by cohort. Incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the local laboratory.

Vital sign measurements and change from baseline will be summarized at each scheduled time point by cohort using descriptive statistics.

Arithmetic mean of parameters from triplicate ECG will be calculated first for each participant at each planned time point. Then summary statistics of ECG test parameters (mean of triplicate) and change from baseline to each post-dose time point will be calculated. Shift tables for ECG test result category change (normal, abnormal, clinically abnormal) from pre-dose to each post-dose time point showing number and percentage of subjects with movement between categories will be presented by treatment group. Frequency and percentage of subjects experiencing potential QTc prolongation (QTcF > 450) will be summarized at each time point by cohort.

#### 12.6 Pharmacodynamic/Activity Data

PD results will be summarized by cohort.

#### 12.7 Immunogenicity Data

Immunogenicity results will be summarized by cohort.

# 12.8 Interim Analysis

No interim analysis is planned. Safety results will be examined for making dose-escalation decisions; no statistical analyses are planned for aiding these dose-escalation decisions.

# 13 DATA QUALITY ASSURANCE

All data will be entered in a validated electronic data capture system using single data entry. Standard procedures (including following data review guidelines, manual clinical review based on subject profiles, computerized validation to produce queries, and maintenance of an audit file which includes all database modifications) will be followed to ensure accurate data. Clinical personnel will review all data listings for outliers, data inconsistencies, and spelling errors.

During the study, a study site monitor will make site visits to review protocol compliance, compare electronic case report forms (eCRFs) against individual subject medical records, assess drug accountability, and ensure that the study is being conducted using pertinent regulatory requirements. eCRF entries will be verified with source documentation. The review of medical records will be performed in a manner to ensure that subject confidentiality is maintained. Checking the eCRFs for completeness, clarity and cross checking with source documents is required to monitor the progress of the study. Direct access to source data is also required for inspections and audits, and will be carried out giving due consideration to data protection and medical confidentiality. Each Investigator will have assured Syntimmune of full access to complete source data for study participants and associated necessary support at all times.

In addition to routine monitoring procedures, audits of clinical research activities in accordance with standard operating procedures (SOPs) may be performed to evaluate compliance with the principles of GCP. A regulatory authority may also wish to conduct an inspection (during the study or even after its completion). If a regulatory authority requests an inspection, the Investigator must immediately inform Syntimmune that this request has been made. Study conduct may be assessed during the study by a Clinical Quality Assurance representative(s) to ensure that the study is conducted in compliance with the protocol. This designee, as well as the site monitor, will be permitted to inspect the study documents (study protocol, eCRFs, investigational product accountability, original study-relevant medical records). All subject data will be treated confidentially. During the clinical study, access will be available to Syntimmune or their designee (e.g., contract research organization [CRO]) to view the eCRFs after completion of the individual sections of the study. Furthermore, the study protocol, each step of the data-recording procedure and the handling of the data as well as the study report may be subject to independent review by a Quality Assurance representative. Clinical site and study audits will be conducted as necessary to assure the validity of the study data.

#### 14 STUDY ADMINISTRATION

# 14.1 Study Administrative Structure

The study administration structure is provided in Table 6.

**Table 6:** Study Administrative Structure



# 14.2 Ethical Conduct of the Study

The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH E6 Tripartite Guideline (January 1997), and in general, be conducted in a manner consistent with the principles described in the Declaration of Helsinki. The Investigator will ensure that the conduct of the study complies with the basic principles of GCP as outlined in the current version of 21 CFR, subpart D, Part 312, "Responsibilities of Sponsors and Investigators", Part 50, "Protection of Human Subjects", and Part 56, "Institutional Review Boards".

#### 14.3 Informed Consent (ICF)

A properly executed, written informed consent document, in compliance with 21 CFR, Part 50 and the ICH guidelines, will be obtained from each subject before the subject is entered into the study and before any study screening procedure is performed that involves risk. Attention will be directed to the basic elements required for incorporation into the informed consent under US Federal Regulations for Protection of Human Subjects (21 CFR 50.25[a]) and (21 CFR 50.25[b]), as necessary.

Sample ICFs will be supplied to each site. Syntimmune or its designee must review any proposed deviations from the sample ICF. The final IRB-approved document must be provided to Syntimmune for regulatory purposes.

It is the responsibility of the Investigator, or a person designated by the Investigator, to obtain written informed consent from each subject (or the subject's legally authorized representative) participating in this study after adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study. In the case where the subject is unable to read, an impartial witness should be present during the entire informed consent discussion. After the subject has orally consented to participation in the trial, the witness' signature on the form will attest that the information in the consent form was accurately explained and understood. A copy of the ICF must be provided to the subject or to the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

The eCRF for this study contains a section for documenting informed subject consent, and this must be completed appropriately. Signed ICFs must remain in each subject's study file and must be available for verification by site monitors at any time. If new safety information results in significant changes in the risk/benefit assessment, the consent form should be reviewed and updated as necessary. All subjects (including those already being treated) should be informed of the new information, should be given a copy of the revised form, and should give their consent to continue in the study.

#### 14.4 Institutional Review Board

This study is being conducted under US IND 128152. This protocol (and any modifications) and appropriate consent procedures must be reviewed and approved by an IRB. This board must operate in accordance with the current federal or local regulations. The Investigator will send a letter or certificate of IRB approval to Syntimmune (or designee) before subject enrollment and whenever subsequent modifications to the protocol are made.

# **14.5** Dose Escalation Committee

The DEC will be responsible for confirming the safety of the investigative product prior to dose escalation, as well as the dose level for each successive cohort. In addition, over the course of the study, the DEC will review any drug-related SAEs to determine if modifications to the study or other measures are necessary to ensure the safety of the subjects. The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To

assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organizations review the data and participate in the discussions.

# 14.6 Future Use of Subject Samples

Not all the tissue and blood components obtained during this study may be required for the tests that are part of the clinical trial. Available samples may be used for additional research. This research will help to understand disease subtypes, drug response and AE, and possibly identify new drug targets or biomarkers that predict subject response to treatment. The use of the samples for internal research will be done using the guidelines defined by the FDA guidance for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individual Identifiable (issued 25 April 2006) and the European Medicines Agency (EMA) Reflection Paper on Pharmacogenetic Samples, Testing and Data Handling (Doc. Ref.

EMEA/CHMP/PGxWP/201914/2006; 15 November 2007). If a subject requests destruction of their tissue and blood samples and the samples have not yet been de-identified, Syntimmune will destroy the samples as described in this FDA guidance. Syntimmune will notify the Investigator in writing that the samples have been destroyed.

#### 15 CONDITIONS FOR MODIFYING THE PROTOCOL

Protocol modifications to ongoing studies must be made only after consultation between a Syntimmune representative and the Investigator. Protocol modifications will be prepared, reviewed, and approved by Syntimmune representatives.

All protocol modifications must be submitted to the IRB for information and approval in accordance with local requirements, and to regulatory agencies if required. Approval must be obtained before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to study subjects, or when the change involves only logistical or administrative aspects of the trial (e.g., change in site monitor, change of telephone number).

# 16 CONDITIONS FOR TERMINATING THE STUDY

Syntimmune has the right to terminate the study at any time. In terminating the study, Syntimmune and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests.

# 17 STUDY DOCUMENTATION, CRFS, AND RECORD KEEPING

# 17.1 Investigator's Files and Retention of Documents

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into 2 separate categories as follows: (1) Investigator's study file and (2) subject clinical source documents.

The Investigator's study file will contain the protocol and protocol amendments, eCRFs, query forms, IRB and governmental approval with correspondence, sample informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

Subject clinical source documents (usually predefined by the project to record key efficacy and safety parameters independent of the eCRFs) may include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, electroencephalogram, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject screening and enrollment logs. The Investigator must keep these 2 categories of documents on file for at least 2 years following the marketing application approval date for the study treatment and for the indication being investigated or for 2 years after the development program is discontinued and the FDA notified. After that period, the documents may be destroyed subject to local regulations with prior written permission from Syntimmune. If the Investigator wants to assign the study records to another party or move them to another location, Syntimmune must be notified in advance.

If the Investigator cannot guarantee the archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and Syntimmune to store these in a sealed container outside of the study site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storing outside of the study site.

# 17.2 Source Documents and Background Data

Investigators must maintain adequate and accurate source documents on which the eCRFs for each subject are based. They are separate and distinct from the eCRFs.

These records include detailed notes on the following:

- Medical history
- Date and time of informed consent with Health Insurance Portability and Accountability
  Act (HIPAA) authorization either contained in the ICF or presented to the subject
  candidate as a standalone document
- Description of the complete consenting process
- The basic identifying information that linked the subject's medical record with the eCRFs
- The results of all diagnostic tests performed, diagnoses made, therapy provided, and any other data on the condition of the subject
- The medical condition of the subject during their involvement in the study
- All AEs
- The subject's exposure to the study medication
- The subject's exposure to any concomitant therapy
- All relevant observations and data on the condition of the subject throughout the trial
- Justification for all entries in the subject's eCRF

A subject log of all potentially eligible subjects considered, but not consented, for obvious deviations from the entry criteria, will be kept at each site. The log will contain subjects' initials, diagnosis, eligibility, or, if not eligible, reason for not consenting. All consented subjects will be logged, regardless of whether they ultimately enroll.

Upon request, the Investigator will supply Syntimmune with any required background data from the study documentation or clinic records. This is particularly important when eCRFs are illegible or when errors in data transcription are suspected. In case of special problems or governmental queries or requests for audit inspections, it is also necessary to have access to the complete study records, provided that subject confidentiality is protected.

#### 17.3 Audits and Inspections

The Investigator should understand that source documents for this study should be made available to appropriately qualified personnel from Syntimmune (or designee), or to health authority inspectors after appropriate notification. The verification of the eCRF data must be by direct inspection of source documents.

# 17.4 Electronic Case Report Forms

Clinical trial data for this study will be captured on eCRF designed for computer processing and analysis. This computerized system will be validated and compliant with 21 CFR Part 11. Corrections to data will be made using 21 CFR Part 11, Electronic Records; Electronic Signatures. If corrections are made after review and sign-off by the Investigator, he/she must be aware of the changes and provide written acknowledgement. There will also be an electronic audit trail. Corrections on paper CRFs must be initialed and dated by the person making the change. The Investigator agrees to provide all information requested on the eCRF in an accurate manner using instructions provided. The Investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported to Syntimmune in the eCRF and in all required reports.

An eCRF is required to be submitted for every subject who receives any amount of study drug. This includes submission of retrievable data on subjects who withdraw before completion of the study. Prior to submission, eCRFs must be reviewed for completeness and accuracy, and signed and dated where either indicated, by the Principal Investigator or authorized delegate from the study staff. If a subject stops treatment or terminates from the study, the dates and reasons must be noted on the eCRF.

#### 18 MONITORING THE STUDY

It is understood that the responsible Syntimmune site monitor (or designee) will contact and visit the Investigator regularly and will be allowed on request to inspect the various records of the trial (eCRFs and other pertinent data) if subject confidentiality is maintained in accordance with local requirements.

It will be the site monitor's responsibility to inspect the eCRFs at regular intervals throughout the study, to verify the adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The site monitor should have access to laboratory test reports and other subject records needed to verify the entries on the eCRF. The Investigator (or designee) must agree to cooperate with the site monitor to ensure that any problems detected during these monitoring visits are resolved.

#### 19 CONFIDENTIALITY OF TRIAL DOCUMENTS AND SUBJECT RECORDS

The Investigator must ensure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On eCRFs or other documents submitted to Syntimmune, subjects should be identified by an identification code and not by their names. The Investigator should keep a subject enrollment log showing codes, names, and addresses. The Investigator should maintain documents not for submission to Syntimmune (e.g., subjects' written consent forms) in strict confidence.

Authorized regulatory officials and Syntimmune personnel (or their representatives) will be allowed full access to inspect and copy the records. All study drugs, subject bodily fluids and tissue, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by Syntimmune.

The Principal Investigator also agrees that all information received from Syntimmune, including but not limited to the IB, this protocol, eCRFs, the INDs, and any other study information remain the sole and exclusive property of Syntimmune during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from the sponsor. The Principal Investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 20 PUBLICATION OF DATA AND PROTECTION OF TRADE SECRETS

The results of this study may be published or presented at scientific meetings. The Investigator agrees that any manuscript or abstract they author may be published only after receiving written permission from Syntimmune.

If Syntimmune coordinates a publication or presentation of study results from all study sites, the participation of Investigator or other representatives of study site as a named author shall be determined in accordance with Syntimmune policy and generally accepted standards for authorship.

#### 21 REFERENCES

Agarwal S, Cunningham-Rundles C. Assessment and clinical interpretation of reduced IgG values. Ann Allergy Asthma Immunol. 2007;99(3):281-283. Epub 2007/10/04.

Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID), which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. Clin Exp Immunol. 2013;174(2):203-211. Epub 2013/07/19.

Bugelski PJ, Treacy G. Predictive power of preclinical studies in animals for the immunogenicity of recombinant therapeutic proteins in humans. Curr Opin Mol Ther. 2004;6(1):10-16. Epub 2004/03/12.

Eming R, Hertl M. Immunoadsorption in pemphigus. Autoimmunity. 2006;39(7):609-616. Epub 2006/11/15.

Furst DE. Serum immunoglobulins and risk of infection: how low can you go? Semin Arthritis Rheum. 2009;39(1):18-29. Epub 2008/07/16.

Gonzalez-Quintela A, Alende R, Gude F, et al. Serum levels of immunoglobulins (IgG, IgA, IgM) in a general adult population and their relationship with alcohol consumption, smoking and common metabolic abnormalities. Clin Exp Immunol. 2008;151(1):42-50. Epub 2007/11/17.

International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) (2011). S6(R1) Preclinical Safety Evaluation of Biotechnology-Derived Pharmaceuticals. Accessed 03 June 2016.

http://www.ich.org/products/guidelines/safety/safety-single/article/preclinical-safety-evaluation-of-biotechnology-derived-pharmaceuticals.html.

Jolliff CR, Cost KM, Stivrins PC, et al. Reference intervals for serum IgG, IgA, IgM, C3, and C4 as determined by rate nephelometry. Clin Chem. 1982;28(1):126-128. Epub 1982/01/01.

Keystone E, Fleischmann R, Emery P, et al. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007;56(12):3896-3908. Epub 2007/12/01.

McMillan SA, Douglas JP, Archbold GP, McCrum EE, Evans AE. Effect of low to moderate levels of smoking and alcohol consumption on serum immunoglobulin concentrations. J Clin Pathol. 1997;50(10):819-822. Epub 1998/02/14.

Nixon AE, Chen J, Sexton DJ, et al. Fully human monoclonal antibody inhibitors of the neonatal fc receptor reduce circulating IgG in non-human primates. Front Immunol. 2015;6:176. Epub 2015/05/09.

Ponce R, Abad L, Amaravadi L, et al. Immunogenicity of biologically-derived therapeutics: assessment and interpretation of nonclinical safety studies. Regul Toxicol Pharmacol. 2009;54(2):164-182. Epub 2009/04/07.

Roopenian DC, Christianson GJ, Sproule TJ, et al. The MHC class I-like IgG receptor controls perinatal IgG transport, IgG homeostasis, and fate of IgG-Fc-coupled drugs. J Immunol. 2003;170(7):3528-3533. Epub 2003/03/21.

Schmaldienst S, Mullner M, Goldammer A, et al. Intravenous immunoglobulin application following immunoadsorption: benefit or risk in patients with autoimmune diseases? Rheumatology. 2001;40(5):513-521. Epub 2001/05/24.

van Vollenhoven RF, Emery P, Bingham CO, 3rd, et al. Long-term safety of rituximab in rheumatoid arthritis: 9.5-year follow-up of the global clinical trial programme with a focus on adverse events of interest in RA patients. Ann Rheum Dis. 2013;72(9):1496-1502. Epub 2012/11/09.

Appendix A: NCI CTCAE, Version 4.03

# Common Terminology Criteria for Adverse Events (CTCAE)

# Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

#### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

# Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

Publish Date: May 28, 2009

#### **Quick Reference**

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

#### **Components and Organization**

#### SOC

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### **CTCAE Terms**

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

#### **Definitions**

A brief definition is provided to clarify the meaning of each AE term.

#### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

#### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

#### Activities of Daily Living (ADL)

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

\*\*Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

<sup>†</sup> CTCAE v4.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).
## CONTENTS

| SOC | Page |
|---|---|
| Blood and lymphatic system disorders | 3 |
| Cardiac disorders | 4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 9 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | <b>7</b> 6 |
| Vascular disorders | <b>7</b> 7 |

| | В | lood and lymphatic system | em disorders | | |
|---|---|---|---|---|---|
| | | | Grade | T | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| nemia | Hemoglobin (Hgb) <lln -="" 10.0="" 100="" 6.2="" <lln="" dl;="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL; &lt;6.2 - 4.9 mmol/L; &lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL; &lt;4.9 mmol/L; &lt;80 g/L; transfusion indicated</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | red by an reduction in the amount on the palpitations of the heart, soft syst | • | • • • | ay include pallor of the skin and m | nucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25% reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50% reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder characteriz | ed by the inability of the bone mar | row to produce hematopoietic ele | ments. | | |
| Disseminated intravascular coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by systemic pathological activa<br>s depleted of platelets and coagula | | which results in clot formation thro | oughout the body. There is an incr | rease in the |
| Febrile neutropenia | - | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>degrees F) for more than one ho | red by an ANC <1000/mm3 and a sour. | single temperature of >38.3 degre | es C (101 degrees F) or a sustaine | ed temperature of >=38 degrees 0 | C (100.4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate widespread erythrocyte ce | Il membrane destruction. | | _ |
| Hemolytic uremic syndrome | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteriz | ed by a form of thrombotic microal | ngiopathy with renal failure, hemo | lytic anemia, and severe thromboo | cytopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of leucostasis; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate an increased number of w | nite blood cells in the blood. | | • |
| _ymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in a lymph node. | | | |
| Spleen disorder | Incidental findings (e.g., Howell-<br>Jolly bodies); mild degree of<br>thrombocytosis and<br>leukocytosis | Prophylactic antibiotics indicated | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder of the splee | en. | | | | |
| Thrombotic thrombocytopenic<br>purpura | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | ed by the presence of microangion | • | cytopenic purpura, fever, renal abr | normalities and neurological abnor | malities suc |
| as seizures, hemiplegia, and visu | ual disturbances. It is an acute or s | subacute condition. | T | T | |
| Blood and lymphatic system disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute coronary syndrome | - | Symptomatic, progressive angina; cardiac enzymes normal; hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | | • | dium secondary to coronary artery | disease. The clinical presentation | covers a |
| | unstable angina to myocardial infa | | | | I |
| Aortic valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in aortic valve func | tion or structure. | T | T | |
| Asystole | Periods of asystole; non-urgent medical management indicated | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia without cardi | ac electrical activity. Typically, this | is accompanied by cessation of the | ne pumping function of the heart. | |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>originates above the ventricles. | ed by a dysrhythmia without disce | rnible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz atria. | ed by a dysrhythmia with organize | ed rhythmic atrial contractions with | a rate of 200-300 beats per minut | e. The rhythm disturbance origina | tes in the |
| Atrioventricular block complete | - | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with complete | e failure of atrial electrical impulse | conduction through the AV node t | o the ventricles. | • |
| Atrioventricular block first<br>degree | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | - | - | - |
| | ed by a dysrhythmia with a delay i<br>interval greater than 200 milliseco | | tion of an electrical impulse throug | gh the atrioventricular (AV) node be | eyond 0. |
| Cardiac arrest | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by cessation of the pumping fu | nction of the heart. | , | | • |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by substernal discomfort due to | o insufficient myocardial oxygenati | on. | | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by pathological irregularities in | the cardiac conduction system. | | | |
| Constrictive pericarditis | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | ı<br>ed by a thickened and fibrotic peri | ।<br>icardial sac; these fibrotic changes | impede normal myocardial function | 1 | ı<br>e action. |
| Definition: A disorder characteriz | , a iibiolio poli | , moss mande ondriges | Severe with symptoms at rest or | Life-threatening consequences; | Death |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic<br>dysfunction | - | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | red by failure of the left ventricle to<br>nea, orthopnea, and other signs ar | | • . | e and in end-diastolic volume. Clin | ical |
| Mitral valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in mitral valve funct | ion or structure. | | | |
| Mobitz (type) II atrioventricular<br>block | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with relatively<br>atrioventricular (AV) node to the ve | · · | block of an atrial impulse. This is t | ne result of intermittent failure of a | trial electric |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a progre<br>on through the atrioventricular (AV) | | ior to the blocking of an atrial impu | lse. This is the result of intermitter | nt failure of |
| Myocardial infarction | - | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences;<br>hemodynamically unstable | Death |
| Definition: A disorder characteriz | ed by gross necrosis of the myoca | rdium; this is due to an interruptio | n of blood supply to the area. | | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characteriz | ed by inflammation of the muscle | tissue of the heart. | | | |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by an unpleasant sensation of | irregular and/or forceful beating of | the heart. | | |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characteriz<br>originates in the atria. | ed by a dysrhythmia with abrupt o | nset and sudden termination of at | rial contractions with a rate of 150- | 250 beats per minute. The rhythm | disturbanc |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by fluid collection within the per | ricardial sac, usually due to inflam | mation. | | |
| Pericardial tamponade | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an increase in intrapericardi | al pressure due to the collection o | f blood or fluid in the pericardium. | | |
| Pericarditis | Asymptomatic, ECG or physical findings (e.g., rub) consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic consequences (e.g., pericardial constriction) | Life-threatening consequences; urgent intervention indicated | Death |
| | • | • | • | • | |

| | 1 | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in pulmonary valve | function or structure. | T | T | 1 |
| Restrictive cardiomyopathy | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | ed by an inability of the ventricles | - | | 1 | |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., ventricular assist device);<br>heart transplant indicated | Death |
| Definition: A disorder characteriz | ed by impairment of right ventricul | ar function associated with low eje | ection fraction and a decrease in n | notility of the right ventricular wall. | 1 |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with alternation | | 1 | 1 | |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical intervention indicated | Severe, medically significant,<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | | that originates in the sinus node. | | |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mir | nute that originates in the sinus no | ode.<br>T | 1 |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mir | nute that originates above the ven | tricles. | 1 |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| | ed by a defect in tricuspid valve fu | | | | |
| Ventricular arrhythmia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia that originate | s in the ventricles. | 1 | 1 | 1 |
| Ventricular fibrillation | - | - | - | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz ventricles. | ed by a dysrhythmia without disce | rnible QRS complexes due to rapi | d repetitive excitation of myocardi | al fibers without coordinated contra | action of the |
| Ventricular tachycardia | - | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mir | nute that originates distal to the bu | indle of His. | |
| Wolff-Parkinson-White<br>syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of an accesso | ry conductive pathway between th | e atria and the ventricles that cau | ses premature ventricular activatio | n. |
| Cardiac disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Congenital, familial and genetic disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Congenital, familial and genetic | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| disorders - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| | | Ear and labyrinth dis | sorders | | |
|---|---|---|---|---|---|
| | | <u> </u> | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the ear. | | | |
| External ear inflammation | External otitis with erythema or dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis; stenosis or osteomyelitis; necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation, swelling and r | edness to the outer ear and ear c | anal. | ' | |
| External ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the external ear region. | • | • | , |
| Hearing impaired | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: subjective change in hearing in the absence of documented hearing loss. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. Pediatric (on a 1, 2, 3, 4, 6 and | least one ear; therapeutic intervention indicated. Adults not enrolled in Monitoring Program: hearing loss with hearing aid or intervention indicated; limiting self care ADL. Pediatric (on a 1, 2, 3, 4, 6 and | Adults: Decrease in hearing to profound bilateral loss (absolute threshold >80 dB HL at 2 kHz and above); non-servicable hearing. Pediatric: Audiologic indication for cochlear implant and additional speech-language related services indicated. | - |
| | shift >20 dB at 8 kHz in at least one ear. | 8 kHz audiogram): Threshold<br>shift >20 dB at 4 kHz and above<br>in at least one ear. | 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids; threshold shift >20 dB at 3 kHz and above in at least one ear; additional speech-language related services indicated. | | |
| Definition: A disorder characteriz | red by partial or complete loss of the | ne ability to detect or understand s | ounds resulting from damage to e | ar structures. | |
| Middle ear inflammation Definition: A disorder characteriz | Serous otitis ted by inflammation (physiologic re | Serous otitis, medical intervention indicated sponse to irritation), swelling and | Mastoiditis; necrosis of canal soft tissue or bone redness to the middle ear. | Life-threatening consequences; urgent intervention indicated | Death |
| Tinnitus | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by noise in the ears, such as rir | nging, buzzing, roaring or clicking. | 1 | T | |
| Vertigo | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz<br>vertigo). | ted by a sensation as if the externa | al world were revolving around the | patient (objective vertigo) or as if | he himself were revolving in space | e (subjective |
| Vestibular disorder | - | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by dizziness, imbalance, nause | ea, and vision problems. | | | |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Endocrine disord | lers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adrenal insufficiency | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rs when the adrenal cortex does not | · | cortisol and in some cases, the ho | ormone aldosterone. It may be due | to a disorde |
| | son's disease or primary adrenal ins | | 0 " " | | |
| Cushingoid | Mild symptoms; intervention not indicated | intervention indicated | Severe symptoms, medical intervention or hospitalization indicated | - | - |
| Definition: A disorder character<br>osteoporosis, usually due to ex | ized by signs and symptoms that re ogenous corticosteroids. | semble Cushing's disease or sync | lrome: buffalo hump obesity, striat | tions, adiposity, hypertension, diab | etes, and |
| Delayed puberty | - | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | - | - |
| Definition: A disorder character | ized by unusually late sexual maturi | ty. | | | |
| Growth accelerated | - | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | - | - |
| Definition: A disorder character | ized by greater growth than expecte | d for age. | | | |
| Hyperparathyroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character the blood). | ized by an increase in production of | parathyroid hormone by the para | thyroid glands. This results in hype | ercalcemia (abnormally high levels | of calcium i |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid suppression therapy indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by excessive levels of thyroid h | ormone in the body. Common car | uses include an overactive thyroid | gland or thyroid hormone overdos | se. |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical intervention or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | | • |
| Hypothyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by a decrease in production of | thyroid hormone by the thyroid gla | and. | 1 | |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical<br>markers of puberty for females<br><8 years and males <9 years | - | - | - |
| Definition: A disorder character<br>9 for boys. | ized by unusually early developmen | t of secondary sexual features; th | e onset of sexual maturation begir | ns usually before age 8 for girls an | d before age |
| √irilization | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | ized by inappropriate masculinization | n occurring in a female or prepub | ertal male. | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Adverse Event 1 2 3 3 4 6 8 Burred Vision Potential control of the control indicated plant of the control of t | | | Eye di | sorders | | |
|---|---|---|---|---|---|---|
| Biurned vision intervention not indicated production of undersided production of undersided production of undersided diagnostic characterized by visual perception of undersided diagnostic characterized by visual perception of undersided diagnostic characterized by visual perception of undersided diagnostic characterized by partial or complete gracely of the cystallities less of one or both eyes. This results in a decrease in visual acuty (wome this 2004) but better but an 20020, perceptive undersided (e.g., artibliotics), limiting self-care ADL. Definition: A disorder characterized by partial or complete gracely of the cystallities less of one or both eyes. This results in a decrease in visual acuty and eventual bindeness of undersided the production of the control of the cystallities less of one or both eyes. This results in a decrease in visual acuty and eventual bindeness of undersided the production of the cystallities less of one or both eyes. This results in a decrease in visual acuty and eventual bindeness of undersided the production of the cystallities less of one or both eyes. This results in a decrease in visual acuty and eventual bindeness of undersided the production of the cystallities less of one or both eyes. This results in a decrease in visual acuty and eventual bindeness of undersided the production of the cystallities less of the cystallities less of the original control of the cystallities less of the | | | | Grade | | |
| Definition: A disorder characterized by visual perception of underest or fuzzy images. Definition: A disorder characterized by visual perception of underest or fuzzy images. Definition: A disorder characterized by partial or correlated operations of understand and under the content of the | Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Appropriate control of disposition for the correction of disposition for the correction of disposition for the correction of the correction of disposition for the correction of disposition of the correction of the correction of disposition of the correction of the corre | | | instrumental ADL | Limiting self care ADL | - | - |
| diagnosts observations only, decrease in visual aculty (2040 or better) (2040 or better) (source than 20200); operative than 20200); operative than 20200); operative than 20200); operative than 20200); operative indicated (e.g., antibodes) (indicated (e.g., antibodes) (e.g., antibodes) (indicated (e.g., antibodes) (e.g | | | | 0 | Dii | |
| Uniterated. Conjunctivitis Asymptomatic or mild symptoms; intervention not indicated (e.g., antibiotics), limiting self care ADL, indicated (e.g., antibiotics), limiting self care ADL, intervention indicated (e.g., antibiotics), limiting self care ADL; intervention indicated (e.g., antibiotics), limiting self care ADL; declining vision (worse than conjunctiva of the eye. Comeal ulcer - Symptomatic, clinical or looking and redeness to the conjunctiva of the eye. Symptomatic clinical or symptomatic clinical or looking and redeness to the conjunctiva of the eye. Definition: A disorder characterized by an area of epithelial issue loss on the surface of the cornea. It is associated with inflammatory cells in the cornea and anterior chamber. Dry eye Asymptomatic, clinical or symptomatic multiple diagnosis observations only; diagnosis conservations only; diagnosis conservations only; diagnosis conservations only; diagnosis conservations only; diagnosis observations only; distributed by diagnosis observations only; instrumental ADL care ADL: disability distributed by diagnosis observations only; instrumental ADL care ADL: disability distributed by diagnosis observations only; instrumental ADL care ADL: disability distributed by diagnosis observations only; instrumental ADL care ADL: disability distributed by diagnosis observations only; instrumental ADL care ADL: distributed characterized by a sudden or brief burst of light. Ficaters Sympt | Cataract | diagnostic observations only; | decrease in visual acuity | decrease in visual acuity<br>(worse than 20/40 but better<br>than 20/200); operative<br>intervention indicated (e.g., | , , | - |
| Symptoms: intervention not indicated (a g., antibioticals; limiting instrumental ADL. Definition: A disorder characterized by inflammation, swelling and redees to the conjunctivar of the eye. | | erized by partial or complete op | pacity of the crystalline lens of o | one or both eyes. This results in | n a decrease in visual acuity an | d eventual blindness if |
| Symptomatic: medical (e.g., Limiting self care ADL: declining vision (worse than to 20/200) affected (20/200 or worse) in the volcal agents; limiting instrumental ADL (20/200 or worse) in the volcal agents; limiting instrumental ADL (20/200 or worse) in the 20/200 or | Conjunctivitis | symptoms; intervention not | intervention indicated (e.g., antibiotics); limiting | Limiting self care ADL | - | - |
| Intervention indicated (e.g., doclaiming vision (worse than a factored cycle) in the appointmental ADL policial agents; limiting instrumental ADL policial for the factor of the cornea. It is associated with inflammatory cells in the cornea and anterior chamber. Dry eye Asymptomatic; clinical or diagnostic observations only, mild symptoms releved by ubricans. Symptomatic; runtiple agents indicated; limiting mild symptoms releved by ubricans. A disorder characterized by dryness of the cornea and conjunctiva. Extraocular muscle paresis Asymptomatic; clinical or diagnostic observations only instrumental ADL pefinition: A disorder characterized by incomplete paralysis of an extraocular muscle. Wild pain Modarta pain; limiting advantage in the cornea and conjunctiva. Severe pain; limiting self care ADL; disabiling assume that ADL pefinition: A disorder characterized by a sensation of marked discomfort in the eye. Severe pain; limiting self care ADL; disabiling assumental ADL pefinition: A disorder characterized by a sensation of marked discomfort in the eye. Severe pain; limiting self care ADL; disabiling assumental ADL pefinition: A disorder characterized by a sudden or brief burst of light. Evalid function disorder Assumentage and the properties of the experimental ADL pefinition: A disorder characterized by a sudden or brief burst of light. Evaluation of the properties of the experimental ADL pefinition: A disorder characterized by a individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Elicope and infected eye in the experimental ADL pefinition: A disorder characterized by an increase in pressure in the eyeball dust to obstruction of the aqueues humor outflow. Evaluation of the aqueues humor outf | Definition: A disorder characte | erized by inflammation, swelling | and redness to the conjunctive | a of the eye. | | |
| Dry eye Asymptomatic; clinical or diagnostic observations only; mild symptoms relieved by furbicants Definition: A disorder characterized by dryness of the comea and conjunctiva. Extraocular muscle paresis Asymptomatic; clinical or diagnostic observations only instrumental ADL Compared the comea and conjunctiva. Extraocular muscle paresis Asymptomatic; clinical or diagnostic observations only of diagnostic observations only of the properties of the comea and conjunctiva. Extraocular muscle paresis Asymptomatic; clinical or diagnostic observations only of the part of diagnostic observations only of the part of the properties of the part of the par | Corneal ulcer | - | intervention indicated (e.g., topical agents); limiting | declining vision (worse than | (20/200 or worse) in the | - |
| diagnostic observations only; bubricants (captured by bubricants) agents indicated; limiting instrumental ADL (captured by bubricants) and conjunctiva. Extraocular muscle parsels Asymptomatic; clinical or diagnostic observations only; bustrumental ADL (captured by diagnostic observations) only; bustrumental ADL (captured by diagnostic observations) only; bustrumental ADL (captured by diagnostic observations) only; bustrumental ADL (captured by diagnostic observations) only; bustrumental ADL (captured by diagnostic observations) only; bustrumental ADL (captured by a sensation of marked discomfort in the eye. Eye pain (captured by a sensation of marked discomfort in the eye. Eyelid function disorder (character/zed by a sensation of marked discomfort in the eye. Eyelid function disorder (character/zed by a sensation of marked discomfort in the eye. Eyelid function disorder (character/zed by impaired eyelid function). Flashing lights (captured by impaired eyelid function). Flashing lights (captured by impaired eyelid function). Floaters (captured by a sudden or brief burst or substrumental ADL (captured by impaired eyelid function). Floaters (captured by a sudden or brief burst or substrumental ADL (captured by a sudden or brief) | Definition: A disorder charact | erized by an area of epithelial ti | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the cornea | and anterior chamber. |
| Extraocular muscle paresis | Dry eye | diagnostic observations only;<br>mild symptoms relieved by | agents indicated; limiting | (<20/40); limiting self care | - | - |
| Definition: A disorder characterized by incomplete paralysis of an extraocular muscle. Eye pain Mild pain Moderate pain; limiting instrumental ADL are ADL care ADL care ADL Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention indicated; limiting instrumental ADL Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting Instrumental ADL Definition: A disorder characterized by an individual seeing sobsets before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. EloP causing early visual field deficits; multiple topical topical agent for intervention; or oral agents indicated; limiting agent care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outllow. Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outllow. Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting instrumental ADL limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outllow. Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting instrumental ADL limiting self care ADL elimiting | Definition: A disorder characte | erized by dryness of the cornea | and conjunctiva. | | | |
| Eye pain Mild pain Moderate pain; limiting instrumental ADL care ADL Care ADL Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated; limiting instrumental ADL limiting self care ADL; operative intervention indicated (limiting instrumental ADL limiting self care ADL Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Care ADL Limiting self care ADL Limiting self care ADL ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL Limiting self care ADL ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit in ovisual field deficit; multiple topical or oral agents indicated; limiting instrumental ADL limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting limiting agents; limiting agents; limiting agents; limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Extraocular muscle paresis | | | | - | - |
| Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated of limiting intervention indicated; limiting self care ADL; operative intervention indicated; limiting self care ADL; operative intervention indicated; limiting performent of indicated operative intervention indicated Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (ElOP) with single topical agent for intervention; no visual field deficit or oral agents indicated; limiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outlow. Keratitis - Symptomatic; medical intervention indicated (e.g., topical agent for a ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL ElioP causing marked visual field deficits (e.g., involving the pressure and inferior visual fields); operative intervention indicated; limiting instrumental ADL Symptomatic; medical intervention indicated (e.g., topical agent of the aqueous humor outlow. Everatitis - Symptomatic out in the eyeball due to obstruction of the aqueous humor outlow. Everation of the aqueous humor outlow. E | Definition: A disorder characte | erized by incomplete paralysis | of an extraocular muscle. | | | T |
| Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated intervention not indicated intervention not indicated; limiting instrumental ADL Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit in visual field deficits; multiple topical agent for intervention; no visual field deficit intervention indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic: medical intervention indicated (e.g., topical agents); limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL - | Eye pain | Mild pain | | | - | - |
| diagnostic observations only, intervention not indicated; limiting instrumental ADL limiting operative intervention indicated limiting instrumental ADL limiting self care ADL | Definition: A disorder characte | erized by a sensation of marked | d discomfort in the eye. | | 1 | |
| Flashing lights Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL | • | diagnostic observations only; intervention not indicated | intervention indicated;<br>limiting instrumental ADL | operative intervention | - | - |
| Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. EloP causing early visual field deficits; multiple topical agent for intervention; no visual field deficit Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Decline in vision (worse than 20/200); limiting self care ADL Declinition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | | | | | | |
| Symptomatic but not limiting ADL Limiting instrumental ADL Limiting self care ADL - Limiting | Flashing lights | | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit witing instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents in the eyeball due to obstruction of the aqueous humor outflow. Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) in the vitreous humor or lens. EIOP causing marked visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Decline in vision (worse than 20/40 but better than 20/200); limiting self care ADL Decline in vision (worse than 20/200 or worse) in the affected eye ADL Definition: A disorder characterized by inflammation to the cornea of the eye. | Definition: A disorder characte | erized by a sudden or brief burs | st of light. | | | |
| Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic but not limiting Symptomatic but not limiting EIOP causing marked visual field deficits (e.g., involving both superior and inferior visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Declinition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Declinition: A disorder characterized by inflammation to the cornea of the eye. EIOP causing marked visual field deficits (e.g., involving both superior and inferior visual fiel | Floaters | | Limiting instrumental ADL | Limiting self care ADL | - | - |
| pressure (EIOP) with single topical agent for intervention; no visual field deficit Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents in visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting 20/40 but better than 20/200); limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Definition: A disorder characte | erized by an individual seeing s | pots before their eyes. The spe | ots are shadows of opaque cell | fragments in the vitreous humo | or or lens. |
| Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Limiting self care ADL Decline in vision (worse than 20/200 or worse) in the affected eye Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Glaucoma | pressure (EIOP) with single topical agent for intervention; | field deficits; multiple topical or oral agents indicated; | field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated; | · ' | - |
| Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Limiting self care ADL Decline in vision (worse than 20/200 or worse) in the affected eye Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Definition: A disorder characte | ·<br>erized by an increase in pressu | re in the eyeball due to obstruc | tion of the aqueous humor out | low. | • |
| Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting | Decline in vision (worse than 20/40 but better than 20/200); limiting self care | Perforation or blindness<br>(20/200 or worse) in the | - |
| | Definition: A disorder characte | erized by inflammation to the co | ornea of the eye. | 1 | Γ | 1 |
| in the another eye | Night blindness | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only | Limiting vision of the affected eye (20/40 or better) | eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| | erized by involvement of the op | · | i | Di: 1 (00/000 ) | |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by swelling around the o | ptic disc. | I | Ι | I |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charact | erized by fear and avoidance of | f light. | 1 | 1 | |
| Retinal detachment | Asymptomatic | Exudative and visual acuity 20/40 or better | Rhegmatogenous or<br>exudative detachment;<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by the separation of the | inner retina layers from the und | derlying pigment epithelium. | | |
| Retinal tear | - | Laser therapy or pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by a small laceration of t | he retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | and floaters. |
| Retinal vascular disorder | - | Topical medication indicated | Intravitreal medication; operative intervention indicated | - | - |
| Definition: A disorder charact | erized by pathological retinal bl | ood vessels that adversely affe | cts vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked<br>decrease in visual acuity<br>(worse than 20/40);<br>disabling; limiting self care<br>ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder involvin | g the retina. | • | | , | • |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better) | Symptomatic, limiting self care ADL; marked decrease in visual acuity (worse than 20/40) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by involvement of the sc | lera of the eye. | T | T | 1 |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | • | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by inflammation to the uv | vea of the eye. | 1 | I . | 1 |
| Vitreous hemorrhage | Asymptomatic or mild symptoms; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by blood extravasation in | nto the vitreous humor. | T | T | T |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | - | - |
| Definition: A disorder of excess | ssive tearing in the eyes; it can | be caused by overproduction of | of tears or impaired drainage of | the tear duct. | 1 |
| Eye disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Sight-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| | erized by swelling of the abdomen. | | <u> </u> | | 1 |
| Abdominal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the abdominal region. | T | | 1 |
| Anal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the opening in the anal | canal to the perianal skin. | | |
| Anal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the anal regio | on. | I | | 1 |
| Anal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the mucous | membrane of the anus. | <del></del> | | |
| Anal necrosis | - | - in the analyzarian | TPN or hospitalization indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by a necrotic process occurring | | Cavara nain, limiting calf care | | |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | erized by a sensation of marked disco | | 0 1 1 1 | | - · |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the anal canal. | | | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammate | ory and necrotic erosive lesion on | the mucosal surface of the anal ca | nal. | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by accumulation of serous or h | emorrhagic fluid in the peritoneal | cavity. | • | |
| Bloating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | - | - | - |
| Definition: A disorder characte | erized by subject-reported feeling of u | uncomfortable fullness of the abdo | men. | | |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the cecum. | | | | |
| Cheilitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | - | - |
| | erized by inflammation of the lip. | T. | 1 | 1 | 1 |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the colon. | 1 | 1 | İ | ı |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an abnormal communication | between the large intestine and | another organ or anatomic site. | | |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the colon. | Т | T | Г | |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | ized by blockage of the normal flow | | | Life in | Б " |
| Colonic perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ized by a rupture in the colonic wall. | | | | 1 |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by a narrowing of the lumen of | the colon. | , | • | • |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by a circumscribed, inflammato | ory and necrotic erosive lesion on t | the mucosal surface of the colon. | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with regular use of laxatives or enemas; limiting instrumental ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by irregular and infrequent or d | ifficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis<br>or periapical abscess or<br>resulting in tooth loss | - | - |
| Definition: A disorder character | ized by the decay of a tooth, in whic | h it becomes softened, discolored | and/or porous. | | |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day<br>over baseline; moderate<br>increase in ostomy output<br>compared to baseline | Increase of >=7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by frequent and watery bowel r | movements. | | | |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment orally; tube feeding or TPN indicated; unstimulated saliva <0.1 ml/min | - | - |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the duodenum and and | other organ or anatomic site. | | 1 |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the duodenur | n. | | 1 | ı |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective operative intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of stomach contents through the | duodenum. | | |
| Duodenal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a rupture in the duodenal w | all. | 1 | 1 | 1 |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the duodenum. | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the duoder | nal wall. | |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| Definition: A disorder characte<br>heartburn, nausea and vomiti | erized by an uncomfortable, often pai | nful feeling in the stomach, resulti | ing from impaired digestion. Sympt | oms include burning stomach, blo | ating, |
| Dysphagia | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely altered eating/swallowing; tube feeding or TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by difficulty in swallowing. | 1 | 1 | 1 | 1 |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent abdominal pain; fever; ileus; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the small ar | nd large intestines. | _ | | |
| Enterovesical fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the urinary bladder and | d the intestine. | | |
| Esophageal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the esophagus and an | other organ or anatomic site. | • | • |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |

| | Gastrointestinal disorders | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by a necrotic process occurring | g in the esophageal wall. | 1 | I | |
| Esophageal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of the contents in the esophagus | | I | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by a sensation of marked disco | omfort in the esophageal region. | 1 | ı | |
| Esophageal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character Esophageal stenosis | ized by a rupture in the wall of the | Symptomatic; altered GI | 0 | 1 15- 41 | Death |
| zsopnagear stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Deam |
| Definition: A disorder character | ized by a narrowing of the lumen of | the esophagus. | | | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by a circumscribed, inflammate | ory and necrotic erosive lesion on | the mucosal surface of the esopha | igeal wall. | |
| Esophageal varices<br>nemorrhage | - | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from esophageal v | varices. | | | |
| Esophagitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered eating/swallowing; oral supplements indicated | Severely altered eating/swallowing; tube feeding, TPN or hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the esopha | geal wall. | | <u> </u> | |
| Fecal incontinence | Occasional use of pads required | | Severe symptoms; elective operative intervention indicated | - | - |
| | ized by inability to control the escap | | | | |
| Flatulence | Mild symptoms; intervention not indicated | psychosocial sequelae | - | - | - |
| | ized by a state of excessive gas in | 1 | 0 1 11 1016 11 | | Ь " |
| Gastric fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by an abnormal communication | n between the stomach and anoth | er organ or anatomic site. | 1 | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the gastric wa | all. | · | | |
| Gastric necrosis | - | - | Inability to aliment adequately by GI tract; radiologic, | Life-threatening consequences; urgent operative intervention | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation | rized by a rupture in the stomach wa | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | | | Caverely altered Cl functions | Life threatening concessions | Dooth |
| Gastric stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the stomach. | | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | rized by a circumscribed, inflammato | ľ | the mucosal surface of the stomac | | 1 |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by inflammation of the stomach | n. | 1 | | |
| Gastroesophageal reflux<br>disease | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | rized by reflux of the gastric and/or d<br>y result in injury to the esophageal m | | , , | nd usually caused by incompetend | e of the lov |
| Gastrointestinal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site. | |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | mfort in the gastrointestinal region | 1. | | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to maintain nutrition with dietary and lifestyle modifications; may need pharmacologic intervention | Weight loss; refractory to medical intervention; unable to maintain nutrition orally | - | - |
| Definition: A disorder characte | rized by an incomplete paralysis of t | he muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small inte | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to aliment orally | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the gingival region. | T | 1 | |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the hemorrho | ids. | 1 | | |
| Hemorrhoids | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characte | rized by the presence of dilated vein | s in the rectum and surrounding a | rea. | | |
| leal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the ileum and another o | organ or anatomic site. | | |
| leal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| | | intervention or minor cauterization indicated | endoscopic, or elective operative intervention indicated | urgent intervention indicated | |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| leal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by blockage of the normal flow | of the intestinal contents in the ile | eum. | 1 | |
| lleal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a rupture in the ileal wall. | | | | |
| lleal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characterize | zed by a narrowing of the lumen of | the ileum. | T | T | |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the ileum. | T | |
| lleus<br>Definition: A disorder characteri: | -<br>zed by failure of the ileum to transp | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Intra-abdominal hemorrhage | | Medical intervention or minor | Transfusion, radiologic, | Life-threatening consequences; | Death |
| mia-asuomina nemormage | | cauterization indicated | endoscopic, or elective operative intervention indicated | urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding in the abdominal c | avity. | _ | | |
| Jejunal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | red by an abnormal communication | n between the jejunum and anoth | er organ or anatomic site. | · | • |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the jejunal wa | all. | 1 | ! | |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents in the je | ejunum. | | |
| Jejunal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ।<br>zed by a rupture in the jejunal wall. | • | | • | • |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a narrowing of the lumen of | the jejunum. | | | |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the jejunun | 1. | |
| _ip pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Lower gastrointestinal | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| hemorrhage | | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | | cauterization indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by bleeding from the lower gas | strointestinal tract (small intestine, | large intestine, and anus). | T | 1 |
| Malabsorption | - | Altered diet; oral intervention indicated | Inability to aliment adequately;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inadequate absorption of nu | trients in the small intestine. Sym | ptoms include abdominal marked | discomfort, bloating and diarrhea. | |
| Mucositis oral | Asymptomatic or mild | Moderate pain; not interfering | Severe pain; interfering with oral | Life-threatening consequences; | Death |
| | symptoms; intervention not | with oral intake; modified diet | intake | urgent intervention indicated | |
| | indicated | indicated | I | | |
| Definition: A disorder characte | erized by inflammation of the oral mu | cosal. | | T | 1 |
| Nausea | Loss of appetite without | Oral intake decreased without | Inadequate oral caloric or fluid | - | - |
| | alteration in eating habits | significant weight loss, | intake; tube feeding, TPN, or | | |
| | | dehydration or malnutrition | hospitalization indicated | | |
| | erized by a queasy sensation and/or | | T | I | I_ |
| Obstruction gastric | Asymptomatic; clinical or | Symptomatic; altered Gl | Hospitalization indicated; | Life-threatening consequences; | Death |
| | diagnostic observations only;<br>intervention not indicated | function; limiting instrumental ADL | elective operative intervention indicated; limiting self care ADL; | urgent operative intervention indicated | |
| | antorvontion not indicated | ,,,,,,, | disabling | maioatou | |
| Definition: A disorder characte | l<br>erized by blockage of the normal flow | of the contents in the stomach | 13 | 1 | I |
| Oral cavity fistula | Asymptomatic; clinical or | | Severely altered GI function; | Life threatening con | Death |
| Oral Cavity IIstula | diagnostic observations only; | Symptomatic; altered GI function | TPN or hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | intervention not indicated | Turiction | elective operative intervention | digent intervention indicated | |
| | | | indicated | | |
| Definition: A disorder characte | erized by an abnormal communication | n between the oral cavity and ano | ther organ or anatomic site. | ! | 1 |
| Oral dysesthesia | Mild discomfort; not interfering | Moderate pain; interfering with | Disabling pain; tube feeding or | _ | _ |
| oran ayooonioona | with oral intake | oral intake | TPN indicated | | |
| Definition: A disorder characte | erized by a burning or tingling sensati | 1 | • | ı | 1 |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| g- | , | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | | cauterization indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by bleeding from the mouth. | • | • | | • |
| Oral pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | _ |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by a sensation of marked disco | mfort in the mouth, tongue or lips | 1 | ! | 1 |
| Pancreatic duct stenosis | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| | diagnostic observations only; | function | tube feeding or hospitalization | urgent operative intervention | Dodui |
| | intervention not indicated | | indicated; elective operative | indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the pancreatic duct. | | | |
| Pancreatic fistula | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| | diagnostic observations only; | function | tube feeding or TPN or | urgent operative intervention | |
| | intervention not indicated | | hospitalization indicated; | indicated | |
| | | | elective operative intervention | | |
| | | | indicated | | |
| Definition: A disorder characte | erized by an abnormal communication | n between the pancreas and anot | ner organ or anatomic site. | 1 | |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| | | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | | cauterization indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by bleeding from the pancreas | | T | T | |
| Pancreatic necrosis | - | - | Tube feeding or TPN indicated; | Life-threatening consequences; | Death |
| | | | radiologic, endoscopic, or | urgent operative intervention | |
| | | | operative intervention indicated | indicated | |
| Definition: A disorder characte | erized by a necrotic process occurring | g in the pancreas. | | | |
| Pancreatitis | - | Enzyme elevation or radiologic | Severe pain; vomiting; medical | Life-threatening consequences; | Death |
| | | findings only | intervention indicated (e.g., | urgent intervention indicated | |
| | | illianigs only | intorvontion indicated (e.g., | argorit intorvormor maioatoa | |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | rized by inflammation of the pancrea | | | | |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or gingivitis; multiple sites of bleeding on probing; moderate bone loss | Spontaneous bleeding; severe bone loss with or without tooth loss; osteonecrosis of maxilla or mandible | - | - |
| Definition: A disorder in the gir | ngival tissue around the teeth. | 1 | | | |
| Peritoneal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | in the peritoneum. | | T | |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the rectum. | | | | |
| Rectal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the rectum and another | r organ or anatomic site. | | |
| Rectal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the rectal wall | and discharged from the anus. | | | |
| Rectal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the mucous | membrane of the rectum. | | | |
| Rectal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | in the rectal wall. | | T | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by blockage of the normal flow | of the intestinal contents in the re | | Г | |
| Rectal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | rized by a sensation of marked disco | | | l . | |
| Rectal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a rupture in the rectal wall. | | | | |
| Rectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the rectum. | | | |
| Rectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function (e.g. altered dietary habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | I | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Retroperitoneal hemorrhage Definition: A disorder characterize | -<br>ted by bleeding from the retroperite | Self-limited; intervention indicated | Transfusion, medical, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Salivary duct inflammation | Slightly thickened saliva; slightly | | Aguta galiyany gland negrasis: | Life threatening concequences: | Death |
| Sanvary duct illiammation | altered taste (e.g., metallic) | Thick, ropy, sticky saliva;<br>markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis;<br>severe secretion-induced<br>symptoms (e.g., thick saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated;<br>limiting self care ADL; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the salivary | duct. | | | |
| Salivary gland fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | n between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe pain; interfering with oral<br>intake; tube feeding, TPN or<br>hospitalization indicated; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the intestinal contents. | | | |
| Small intestinal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the small intesti | ne wall. | | | |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the small intestine. | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on t | the mucosal surface of the small in | testine. | |
| Stomach pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | omfort in the stomach. | 1 | | |
| Γooth development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with oral surgery | Maldevelopment with impairment not surgically correctable; disabling | - | - |
| Definition: A disorder characteriz | ed by a pathological process of the | e teeth occurring during tooth deve | elopment. | | |
| Tooth discoloration | Surface stains | - | - | - | - |
| Definition: A disorder characteriz | red by a change in tooth hue or tint | i. | 1 | | |
| Toothache | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | l <u>-</u> | l - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Typhlitis | - | - | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal signs | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the cecum. | • | • | • | |
| Upper gastrointestinal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the upper gas | trointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | |
| Vomiting | 1 - 2 episodes (separated by 5 minutes) in 24 hrs | 3 - 5 episodes (separated by 5 minutes) in 24 hrs | >=6 episodes (separated by 5<br>minutes) in 24 hrs; tube feeding,<br>TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the reflexive act of ejecting t | he contents of the stomach throuç | h the mouth. | • | • |
| Gastrointestinal disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold;<br>shivering; chattering of teeth | Moderate tremor of the entire body; narcotics indicated | Severe or prolonged, not responsive to narcotics | - | - |
| Definition: A disorder charac | sterized by a sensation of cold that ofte | 1 | 1 ' | I | 1 |
| Death neonatal | - | - | - | - | Death |
| Definition: A disorder charac | terized by cessation of life occurring de | uring the first 28 days of life. | | | |
| Death NOS | - | - | - | - | Death |
| Definition: A cessation of life | that cannot be attributed to a CTCAE | term associated with Grade 5. | | | |
| Edema face | Localized facial edema | Moderate localized facial edema; limiting instrumental ADL | Severe swelling; limiting self care ADL | - | - |
| Definition: A disorder charac | terized by swelling due to excessive flu | uid accumulation in facial tissues. | 1 | | |
| Edema limbs | 5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection | >10 - 30% inter-limb discrepancy in volume or circumference at point of greatest visible difference; readily apparent obscuration of anatomic architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour; limiting instrumental ADL | >30% inter-limb discrepancy in<br>volume; gross deviation from<br>normal anatomic contour;<br>limiting self care ADL | - | - |
| Definition: A disorder charac | terized by swelling due to excessive flu | uid accumulation in the upper or lo | wer extremities. | | |
| Edema trunk | Swelling or obscuration of anatomic architecture on close inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | Gross deviation from normal anatomic contour; limiting self care ADL | - | - |
| Definition: A disorder character Facial pain | terized by swelling due to excessive flu | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |
| Definition: A disorder charac | l<br>sterized by a sensation of marked disco | 1 | INDE | I | I |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest; | Fatigue not relieved by rest, limiting self care ADL | - | - |
| Definition: A disorder charac | terized by a state of generalized weak | ness with a pronounced inability to | summon sufficient energy to acc | omplish daily activities. | |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>104.0 degrees F) for <=24 hrs | >40.0 degrees C (>104.0 degrees F) for >24 hrs | Death |
| Definition: A disorder charac | eterized by elevation of the body's temp | perature above the upper limit of n | ormal. | 1 | |
| Flu like symptoms | Mild flu-like symptoms present | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder charac cough. | sterized by a group of symptoms simila | r to those observed in patients with | n the flu. It includes fever, chills, b | ody aches, malaise, loss of appeti | ite and dry |
| Gait disturbance | Mild change in gait (e.g., wide-<br>based, limping or hobbling) | Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL | Disabling; limiting self care ADL | - | - |
| | eterized by walking difficulties. | 05 - 00 0 - 05 | 20 - 20 | 1-00 d C 00 4 1 | D " |
| Hypothermia | - | 35 - >32 degrees C; 95 - >89.6 degrees F | 32 - >28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C; 82.4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>hypotension, pulmonary edema,<br>acidemia, ventricular fibrillation) | Death |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Infusion related reaction | Mild transient reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by adverse reaction to the infus | ,<br>sion of pharmacological or biologic | cal substances. | • | • |
| Infusion site extravasation | - | Erythema with associated symptoms (e.g., edema, pain, induration, phlebitis) | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by leakage of a pharmacologic<br>sation and marked discomfort at the | • | nfusion site into the surrounding ti | ssue. Signs and symptoms include | e induratio |
| Injection site reaction | Tenderness with or without associated symptoms (e.g., warmth, erythema, itching) | Pain; lipodystrophy; edema; phlebitis | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an intense adverse reaction | i i i i | at the site of an injection. | I | |
| Irritability | Mild; easily consolable | Moderate; limiting instrumental ADL; increased attention indicated | Severe abnormal or excessive response; limiting self care ADL; inconsolable | - | - |
| Definition: A disorder characteriz condition. | zed by an abnormal responsivenes | s to stimuli or physiological arousa | al; may be in response to pain, frig | ht, a drug, an emotional situation | or a medi |
| Localized edema | Localized to dependent areas, no disability or functional impairment | Moderate localized edema and intervention indicated; limiting instrumental ADL | Severe localized edema and intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by swelling due to excessive flu | uid accumulation at a specific anal | tomic site. | T | |
| Malaise | Uneasiness or lack of well being | Uneasiness or lack of well being; limiting instrumental ADL | - | - | - |
| Definition: A disorder characteriz | zed by a feeling of general discomf | ort or uneasiness, an out-of-sorts | feeling. | | |
| Multi-organ failure | - | - | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | Life-threatening consequences<br>(e.g., vasopressor dependent<br>and oliguric or anuric or<br>ischemic colitis or lactic<br>acidosis) | Death |
| Definition: A disorder characteriz | zed by progressive deterioration of | the lungs, liver, kidney and clotting | g mechanisms. | | |
| Neck edema | Asymptomatic localized neck edema | Moderate neck edema; slight<br>obliteration of anatomic<br>landmarks; limiting instrumental<br>ADL | Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by swelling due to an accumula | ation of excessive fluid in the neck | T | T | |
| Non-cardiac chest pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by discomfort in the chest unre | lated to a heart disorder. | | | • |
| Pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | l<br>zed by the sensation of marked dis | ı | j | I | |
| Sudden death NOS | - | - | - | - | Death |
| Definition: An unexpected cessa | tion of life that cannot be attributed | to a CTCAE term associated with | Grade 5. | | |
| General disorders and administration site conditions - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| | | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bile duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Severely altered GI function;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by a narrowing of the lumen of | the bile duct. | 1 | | |
| Biliary fistula | - | Symptomatic and intervention not indicated | Severely altered GI function;<br>TPN indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between the bile ducts and anoth | ner organ or anatomic site. | T | |
| Cholecystitis | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by inflammation involving the g | allbladder. It may be associated w | vith the presence of gallstones. | i | |
| Gallbladder fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Symptomatic or severely altered<br>GI function; TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between the gallbladder and and | other organ or anatomic site. | | |
| Gallbladder necrosis | - | - | - | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | g in the gallbladder. | T | r | |
| Gallbladder obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | zed by blockage of the normal flow | | | | |
| Gallbladder pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the gallbladder region. | | | |
| Gallbladder perforation | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a rupture in the gallbladder ( | waii.<br> - | Asterixis; mild encephalopathy; limiting self care ADL | Moderate to severe encephalopathy; coma; life-threatening consequences | Death |
| | zed by the inability of the liver to me | etabolize chemicals in the body. L | aboratory test results reveal abnor | mal plasma levels of ammonia, bi | lirubin, lac |
| dehydrogenase, and alkaline ph | T | 0 | T | 1 15- 41 | D" |
| Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the liver. | | | | |
| Hepatic necrosis | - | - | - | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the hepatic parenchyma. | _ | | |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the liver region. | 1 | <u> </u> | |
| Perforation bile duct | - | - | Radiologic, endoscopic or elective operative intervention | Life-threatening consequences; urgent operative intervention | Death |

| Hepatobiliary disorders | | | | |
|---|---|---|---|---|
| Grade | | | | |
| 1 | 2 | 3 | 4 | 5 |
| - | Decreased portal vein flow | Reversal/retrograde portal vein flow; associated with varices and/or ascites | Life-threatening consequences; urgent intervention indicated | Death |
| ed by an increase in blood pressur | re in the portal venous system. | | | |
| - | Intervention not indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| ed by the formation of a thrombus | (blood clot) in the portal vein. | | | |
| Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by the formation of a thrombus<br>Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention | Decreased portal vein flow d by an increase in blood pressure in the portal venous system. Intervention not indicated d by the formation of a thrombus (blood clot) in the portal vein. Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention indicated; limiting age- | The symptomatic or mild symptoms; clinical or not indicated The symptoms of indicated or noninvasive intervention indicated in | The content of a thrombus (blood clot) in the portal vein. Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated appropriate instrumental ADL in the content of the conte |

| | | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug<br>fever <38 degrees C (<100.4<br>degrees F); intervention not<br>indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; urgent intervention indicated | Death |
| | ted by an adverse local or general | response from exposure to an alle | | | 1 |
| Anaphylaxis | - | - | Symptomatic bronchospasm,<br>with or without urticaria;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an acute inflammatory react resents with breathing difficulty, dia | | | | ypersensitivit |
| Autoimmune disorder | Asymptomatic; serologic or<br>other evidence of autoimmune<br>reaction, with normal organ<br>function; intervention not<br>indicated | Evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder resulting fratissue constituents. | om loss of function or tissue destru | uction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individ | ual to his owr |
| Cytokine release syndrome | Mild reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | following initial improvement;<br>hospitalization indicated for<br>clinical sequelae (e.g., renal<br>impairment, pulmonary<br>infiltrates) | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| Definition: A disorder characteriz | ed by nausea, headache, tachyca | rdia, hypotension, rash, and short | ness of breath; it is caused by the | release of cytokines from the cells | S. |
| Serum sickness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash, urticaria, antihistamines indicated | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV<br>fluids indicated | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| | ed by a delayed-type hypersensitive foreign antigen. Symptoms include | | | | |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the abdominal cavity. | 1 | 1 | |
| Anorectal infection | Localized; local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | ving the anal area and the rectum. | N/4ibi-4i4if1 | l :f- thti | D#- |
| Appendicitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by acute inflammation to the v | rermiform appendix caused by a pa | athogenic agent. | | |
| Appendicitis perforated | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by acute inflammation to the viceal wall rupture causes the releas | | | | tne |
| Arteritis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving an artery. | T | 1 | |
| Biliary tract infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the biliary tract. | | | |
| Bladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bladder. | | | |
| Bone infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | | | | |
| Breast infection | | Local infection with moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | Severe infection; axillary<br>adenitis; IV antibacterial,<br>antifungal, or antiviral<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Bronchial infection | rized by an infectious process invol | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life threatening consequences: | Death |
| BIOTICIIAI IIIIECUOTI | - | intervention indicated (e.g., antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bronchi. | 1 | 1 | |
| Catheter related infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process that | arises secondary to catheter use. | | | |
| Cecal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | ed by an infectious process involv | | | · · | |
| Cervicitis infection | ed by an infectious process involv | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Del vicius il liection | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | Death |
| | | antifungal, or antiviral) | radiologic or operative | g | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing the uterine cervix. | | | |
| Conjunctivitis infective | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing the conjunctiva. Clinical manif | estations include pink or red color | in the eyes. | |
| Corneal infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characterize | l ed by an infectious process involv | I<br>ing the cornea | | I | I |
| Cranial nerve infection | ca by an infectious process involv | ing the comea. | IV antibiotic antifuncal as | Life threatening assessment | Death |
| Craniai nerve infection | - | - | IV antibiotic, antifungal, or antiviral intervention indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | radiologic or operative | argoni interventien indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing a cranial nerve. | ' | ' | • |
| Device related infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing the use of a medical device. | | | |
| Duodenal infection | - | Moderate symptoms; medical | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., oral | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotics) | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing the duodenum. | T | T | |
| Encephalitis infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | severe changes in mental | | |
| | | | status; self-limited seizure activity; focal neurologic | | |
| | | | abnormalities | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing the brain tissue. | ı | 1 | |
| Encephalomyelitis infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | ed by an infectious process involv | ing the brain and spinal cord tissu | es. | | |
| Endocarditis infective | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| efinition: A disorder characterize | ed by an infectious process involv | ing the endocardial layer of the he | art. | | |
| Committeen: 71 discrete characteriza | | | | | |
| Endophthalmitis | - | Local intervention indicated | Systemic intervention or | Blindness (20/200 or worse) | - |

| | | Infections and infes | | | |
|---|---|---|---|---|---|
| | | T. | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Enterocolitis infectious | - | Passage of >3 unformed stools<br>per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal<br>pain | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated;<br>profuse watery diarrhea with | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the small and large intestines. | signs of hypovolemia; bloody<br>diarrhea; fever; severe<br>abdominal pain; hospitalization<br>indicated | | |
| Esophageal infection | - | Local intervention indicated (e.g., oral antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the esophagus. | | | |
| Eye infection | - Tool by an infectious process involves | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated;<br>enucleation | Death |
| Gallbladder infection | zed by an infectious process involv | ing the eye. | IV antibiotic antifungal or | Life-threatening consequences; | Death |
| Gailbladder iffiection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | urgent intervention indicated | Deam |
| Definition: A disorder characteri | zed by an infectious process involv | ing the gallbladder. | T | T | |
| Gum infection | Local therapy indicated (swish and swallow) | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ring the gums. | • | • | |
| Hepatic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the liver. | | • | |
| Hepatitis viral | Asymptomatic, treatment not indicated | - | Symptomatic liver dysfunction;<br>fibrosis by biopsy; compensated<br>cirrhosis; reactivation of chronic<br>hepatitis | Decompensated liver function<br>(e.g., ascites, coagulopathy,<br>encephalopathy, coma) | Death |
| Definition: A disorder characteri | zed by a viral pathologic process in | nvolving the liver parenchyma. | 1 | | |
| Infective myositis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing the skeletal muscles. | | | |
| Joint infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); needle aspiration indicated (single or multiple) | Arthroscopic intervention indicated (e.g., drainage) or arthrotomy (e.g., open surgical drainage) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process involv | ing a joint. | T | Г | |
| Kidney infection | - | - | IV antibiotic, antifungal, or antiviral intervention indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | T. | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an inflammatory process in | nvolving the larynx. | 1 | 1 | 1 |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characte | rized by an infectious process invol | ving the lips. | | | |
| Lung infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | T | T | I | |
| Lymph gland infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the lymph nodes. | T | T | |
| Mediastinal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the mediastinum. | | | |
| Meningitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by acute inflammation of the r | neninges of the brain and/or spinal | cord. | ' | • |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving a mucosal surface. | | | • |
| Nail infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characte | rized by an infectious process invol | T | | | |
| Otitis externa | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol<br>ptoms include fullness, itching, swe | • | • | ive water exposure (swimmer's ea | r infectior |
| Otitis media | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the middle ear. | | | |
| Ovarian infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | 1 | 1 | Intervention indicated | 1 | 1 |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an infectious process involv | ing the pancreas. | | | |
| Papulopustular rash | Papules and/or pustules<br>covering <10% BSA, which may<br>or may not be associated with<br>symptoms of pruritus or<br>tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | rized by an eruption consisting of pa | | | | p, and upper |
| Paronychia | is rash does not present with whiteh Nail fold edema or erythema; disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical intervention or IV antibiotics indicated; limiting self care ADL | - | - |
| Definition: A disorder character | rized by an infectious process involv | ing the soft tissues around the nai | l. | | |
| Pelvic infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an infectious process involv | ing the pelvic cavity. | T | T | |
| Penile infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an infectious process involv | ing the penis. | | | |
| Periorbital infection | rized by an infectious process involv | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Peripheral nerve infection | lized by an infectious process involv | Localized; local intervention | IV antibiotic antifundal or | Life threatening consequences: | Death |
| | | indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process involv | ing the peripheral nerves. | N/ Albirdia Alf | 1 15- 41 | D# |
| Peritoneal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process involv | | I | I | |
| Pharyngitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by inflammation of the throat. | | | | |
| Phlebitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infest | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize of the infected vein. | ed by an infectious process involvi | ing the vein. Clinical manifestation | s include erythema, marked disco | mfort, swelling, and induration alo | ng the course |
| Pleural infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an infectious process involvi | 1 | N/4!L:-4:4:E1 | 1 15- 41 | D#- |
| Prostate infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the prostate gland. | | | |
| Rash pustular | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characterize | ed by a circumscribed and elevate | d skin lesion filled with pus. | | | |
| Rhinitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | - | - | - |
| | ed by an infectious process involvi | | T | T | |
| Salivary gland infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the salivary gland. | | | |
| Scrotal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the scrotum. | <u> </u> | <u> </u> | |
| Sepsis | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by the presence of pathogenic | microorganisms in the blood strea | m that cause a rapidly progressing | g systemic reaction that may lead | to shock. |
| Sinusitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the mucous membranes of the | paranasal sinuses. | | |
| Skin infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the skin. | I | I | |
| Small intestine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an infectious process involvi | ing the small intestine. | T | T | |
| Soft tissue infection | od by an infestions are seen in | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an infectious process involvi | ing soπ tissues. | n, eg. e | | D " |
| Splenic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | red by an infectious process involv | ing the spleen. | 1 | 1 | |
| Stoma site infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | red by an infectious process involv | ing a stoma (surgically created op | ening on the surface of the body). | 1 | |
| Footh infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing a tooth. | | | |
| Tracheitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing the trachea. | T | I | |
| Upper respiratory infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing the upper respiratory tract (no | se, paranasal sinuses, pharynx, la | rynx, or trachea). | |
| Urethral infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involv | ing the urethra. | | | |
| Urinary tract infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the urinary tract, most commo | nly the bladder and the urethra. | | |
| Uterine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing the endometrium. It may exter | d to the myometrium and parame | trial tissues. | |
| Vaginal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing the vagina. | | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing the vulva. | | | |
| Nound infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an infectious process involv | ing the wound. | I | 1 | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Injury, poisoning and procedural complications Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention | Limiting instrumental ADL; | Limiting self care ADL; elective | 4 | 3 |
| | indicated | operative intervention indicated | surgery indicated | | ļ |
| Definition: A finding of damage affected leg and foot. | to the ankle joint characterized by a | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | y moving the |
| Aortic injury | _ | _ | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| · | | | care ADL; disabling; repair or | evidence of end organ damage; | |
| | | | revision indicated | urgent operative intervention | |
| | | | | indicated | |
| Definition: A finding of damage | | | | | |
| Arterial injury | Asymptomatic diagnostic | Symptomatic (e.g., | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | finding; intervention not indicated | claudication); repair or revision not indicated | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention | |
| | ilidicated | not indicated | Tevision indicated | indicated | |
| Definition: A finding of damage | to an artery. | 1 | | 1 | |
| Biliary anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage | of bile due to breakdown of a biliary | anastomosis (surgical connection | n of two separate anatomic structu | res). | |
| Bladder anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| Definition, A finding of lookage | not indicated | | intervention indicated | indicated | I |
| | of urine due to breakdown of a blad | Generalized | tion of two separate anatomic stru | ctures). | |
| Bruising | area | Generalized | - | - | - |
| Definition: A finding of injury of | the soft tissues or bone characterize | ed by leakage of blood into surrou | nding tissues. | | |
| Burn | Minimal symptoms; intervention | Medical intervention; minimal | Moderate to major debridement | Life-threatening consequences | Death |
| | not indicated | debridement indicated | or reconstruction indicated | | |
| | integrity to the anatomic site of an | | | nicals, direct heat, electricity, flam | es and |
| | e depends on the length and intensi | | | | |
| Dermatitis radiation | Faint erythema or dry desquamation | Moderate to brisk erythema; patchy moist desquamation, | Moist desquamation in areas other than skin folds and | Life-threatening consequences;<br>skin necrosis or ulceration of full | Death |
| | desquamation | mostly confined to skin folds | creases; bleeding induced by | thickness dermis; spontaneous | |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin | |
| | | | | graft indicated | |
| Definition: A finding of cutaneou | us inflammatory reaction occurring a | as a result of exposure to biologica | ally effective levels of ionizing radia | ation. | |
| Esophageal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| D-6-iti | not indicated | | intervention indicated | indicated | l |
| | due to breakdown of an esophagea | | | res). | |
| Fall | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding of sudden r | ा<br>novement downward, usually result | 1 | ı | I | 1 |
| Fallopian tube anastomotic leak | | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| ' | diagnostic observations only; | intervention indicated | endoscopic or elective operative | | |
| | intervention not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage | due to breakdown of a fallopian tub | e anastomosis (surgical connection | on of two separate anatomic structu | ıres). | |
| Fallopian tube perforation | Asymptomatic diagnostic | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| | observations only; intervention | not indicated | operative intervention indicated | urgent operative intervention | |
| Definition: A finding of much | not indicated | | I | indicated (e.g., organ resection) | 1 |
| Definition: A finding of rupture of | <u>'</u> | Communication built are 12 to 1 | Covers over to an all the | Life threater: | Do-#- |
| Fracture | Asymptomatic; clinical or diagnostic observations only; | Symptomatic but non-displaced; immobilization indicated | Severe symptoms; displaced or open wound with bone | Life-threatening consequences; urgent intervention indicated | Death |
| | intervention not indicated | Tobiiization indicated | exposure; disabling; operative | a. gont into vondon indicated | |
| | | | intervention indicated | | |
| S 5 111 A 5 11 A 5 11 A 5 | injury to the bone in which the con | tinuity of the hone is broken | | | |

| | ,, | , poisoning and procedu | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | | Death |
| Gastric ariastorriotic leak | observations only; intervention | intervention indicated | endoscopic or elective operative | Life-threatening consequences; urgent operative intervention | Dealli |
| | not indicated | intervention indicated | intervention indicated | indicated | |
| Definition: A finding of lookens d | ı | tomonic (curried connection of to | • | | 1 |
| | | tomosis (surgical connection of tw | | I | I |
| Gastrointestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| leak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | l |
| Definition: A finding of leakage d | ue to breakdown of a gastrointesti<br>T | nal anastomosis (surgical connec | tion of two separate anatomic struc | ctures). | |
| Gastrointestinal stoma necrosis | - | Superficial necrosis; | Severe symptoms; | Life-threatening consequences; | Death |
| | | intervention not indicated | hospitalization or elective | urgent intervention indicated | |
| | | | operative intervention indicated | | |
| Definition: A finding of a necrotic | process occurring in the gastroint | estinal tract stoma. | | | |
| Hip fracture | - | Hairline fracture; mild pain; | Severe pain; hospitalization or | Life-threatening consequences; | - |
| | | limiting instrumental ADL; non- | intervention indicated for pain | symptoms associated with | |
| | | surgical intervention indicated | control (e.g., traction); operative | neurovascular compromise | |
| | | | intervention indicated | | |
| Definition: A finding of traumatic | injury to the hip in which the contin | nuity of either the femoral head, fe | moral neck, intertrochanteric or su | btrochanteric regions is broken. | |
| Injury to carotid artery | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| , , | | | care ADL (e.g., transient | urgent intervention indicated | |
| | | | cerebral ischemia); repair or | _ | |
| | | | revision indicated | | |
| Definition: A finding of damage to | the carotid artery. | | | • | |
| Injury to inferior vena cava | | _ | _ | Life-threatening consequences; | Death |
| ngary to intener rona cara | | | | urgent intervention indicated | Dou |
| Definition: A finding of demage to | the inferior years sour | 1 | 1 | 13 | ı |
| Definition: A finding of damage to | The interior veria cava. | | | | |
| Injury to jugular vein | - | - | Symptomatic limiting self care | Life-threatening consequences; | Death |
| | | | ADL; disabling; repair or | urgent intervention indicated | |
| | I | I | revision indicated | I | l |
| Definition: A finding of damage to | the jugular vein. | 1 | | | 1 |
| Injury to superior vena cava | Asymptomatic diagnostic | Symptomatic; repair or revision | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | finding; intervention not | not indicated | care ADL; disabling; repair or | evidence of end organ damage; | |
| | indicated | | revision indicated | urgent operative intervention | |
| | | | | indicated | |
| Definition: A finding of damage to | the superior vena cava. | | | | |
| Intestinal stoma leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage of | f contents from an intestinal stoma | (surgically created opening on th | e surface of the body). | | |
| Intestinal stoma obstruction | - | Self-limited; intervention not | Severe symptoms; IV fluids, | Life-threatening consequences; | Death |
| | | indicated | tube feeding, or TPN indicated | urgent operative intervention | |
| | | | >=24 hrs; elective operative | indicated | |
| | | | intervention indicated | | |
| Definition: A finding of blockage | of the normal flow of the contents | of the intestinal stoma. | • | • | • |
| Intestinal stoma site bleeding | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| | clinical exam; intervention not | intervention indicated | indicated; radiologic or | urgent intervention indicated | 20aur |
| | indicated | | endoscopic intervention | a.g.s.ik intorvontion indicated | |
| | | | indicated | | |
| Definition: A finding of blood leak | age from the intestinal stoma | I | ı | I | 1 |
| | | Dertiel reserving of 1 | Complete #ti | Life threatering | De -" |
| Intraoperative arterial injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| | organ/structure indicated | organ/structure indicated | reconstruction of injured | urgent intervention indicated | |
| | | | organ/structure indicated; | | |
| · | 1 | | disabling | I | I |
| Definition: A finding of damage to | o an artery during a surgical proce | dure. | | <u> </u> | |
| Intraoperative breast injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| | organ/structure indicated | organ/structure indicated | reconstruction of injured | urgent intervention indicated | |
| | | | i . | i e | |
| | | | organ/structure indicated; disabling | | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | o the breast parenchyma during a | | , , | 4 | ] 3 |
| Intraoperative cardiac injury | - | - | Primary repair of injured organ/structure indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the heart during a surgical proce | dure. | | | |
| Intraoperative ear injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection of injured organ/structure indicated; disabling (e.g., impaired hearing; impaired balance) | Life-threatening consequences; urgent intervention indicated | Death |
| | o the ear during a surgical procedu | | 1 | T | I |
| Intraoperative endocrine injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the endocrine gland during a sur | gical procedure. | | | |
| Intraoperative gastrointestinal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the gastrointestinal system durin | g a surgical procedure. | | | |
| Intraoperative head and neck<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the head and neck during a surg | ical procedure. | | | |
| Intraoperative hemorrhage | - | - | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical proc | edure. | • | • | • |
| Intraoperative hepatobiliary<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the hepatic parenchyma and/or l | oiliary tract during a surgical pro | cedure. | | |
| Intraoperative musculoskeletal<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the musculoskeletal system duri | ng a surgical procedure. | | | |
| Intraoperative neurological injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Intraoperative ocular injury | o the nervous system during a sur<br>Primary repair of injured | | Complete resection or | l ife threatening consequences | Death |
| muaoperauve oculai injury | organ/structure indicated | Partial resection of injured organ/structure indicated | reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the eye during a surgical proced | ure. | | | |
| Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the kidney during a surgical proc | edure. | | | |
| Intraoperative reproductive tract injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured | Life-threatening consequences; urgent intervention indicated | Death |

| Grade | | | | | | | |
|---|---|---|---|---|---|--|--|
| Adverse Event | 1 | 2 | 3 | 4 | 5 | | |
| | the reproductive organs during a | | • | | | | |
| Intraoperative respiratory injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death | | |
| Definition: A finding of damage to | ।<br>o the respiratory system during a s | urgical procedure. | | ı | 1 | | |
| Intraoperative skin injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death | | |
| Definition: A finding of damage to | the skin during a surgical proced | ure. | | | | | |
| Intraoperative splenic injury | - | Primary repair of injured organ/structure indicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death | | |
| | the spleen during a surgical proc | | 0 11 " | Life iii | L | | |
| Intraoperative urinary injury Definition: A finding of damage to | Primary repair of injured organ/structure indicated the urinary system during a surg | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death | | |
| | Primary repair of injured | Partial resection of injured | Complete resection or | Life threatening consequences: | Death | | |
| Intraoperative venous injury | organ/structure indicated | organ/structure indicated | reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death | | |
| Definition: A finding of damage to | a vein during a surgical procedu | re. | | | | | |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death | | |
| Definition: A finding of leakage of | urine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | | | |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death | | |
| Definition: A finding of leakage du | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | | | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death | | |
| Definition: A finding of leakage du | ue to breakdown of a pancreatic a | nastomosis (surgical connection o | f two separate anatomic structures | s). | | | |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | indicated | Death | | |
| | | anastomosis (surgical connection | | T . | | | |
| Postoperative hemorrhage | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; radiologic, endoscopic, or operative intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death | | |
| | ccurring after a surgical procedur | | F. 4. 4 - 4 - 4 > 70 h | Life the second of | D-: " | | |
| Postoperative thoracic procedure complication | - | Extubated within 24 - 72 hrs postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death | | |
| Definition: A finding of a previous | ly undocumented problem that oc | curs after a thoracic procedure. | | | | | |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental | Severe symptoms; elective operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death | | |
| | mjury, | , poisoning and procedu | • | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | of the intestinal stoma (surgically | | | | |
| Prolapse of urostomy | Asymptomatic; clinical or | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective | Life-threatening consequences; | Death |
| | diagnostic observations only;<br>intervention not indicated | Thirlor revision indicated | operative intervention or major stomal revision indicated | urgent intervention indicated | |
| Definition: A finding of displacem | 1 | | Storriar revision indicated | | l |
| | 1 | NA - d 4 - 4 - 1 44 | NA-i-A di i | 1 : - 4 4 : | D#- |
| Radiation recall reaction<br>(dermatologic) | Faint erythema or dry desquamation | Moderate to brisk erythema; | Moist desquamation in areas other than skin folds and | Life-threatening consequences;<br>skin necrosis or ulceration of full | Death |
| (dernatologic) | desquarration | patchy moist desquamation,<br>mostly confined to skin folds | creases; bleeding induced by | thickness dermis; spontaneous | |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin | |
| | | | | graft indicated | |
| Definition: A finding of acute skin | inflammatory reaction caused by | '<br>drugs, especially chemotherapeut | ic agents, for weeks or months fol | owing radiotherapy. The inflamma | tory react |
| - | liated skin and the symptoms disa | | - | ., | • |
| Rectal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage du | ue to breakdown of a rectal anasto | omosis (surgical connection of two | separate anatomic structures). | | |
| Seroma | Asymptomatic; clinical or | Symptomatic; simple aspiration | Symptomatic, elective radiologic | - | - |
| | diagnostic observations only; | indicated | or operative intervention | | |
| | intervention not indicated | | indicated | | |
| Definition: A finding of tumor-like | collection of serum in the tissues. | | | | |
| Small intestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| leak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage du | ue to breakdown of an anastomosi | is (surgical connection of two sepa | arate anatomic structures) in the si | mall bowel. | |
| Spermatic cord anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| eak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage du | ue to breakdown of a spermatic co | rd anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Spinal fracture | Mild back pain; nonprescription | Moderate back pain; | Severe back pain; | Life-threatening consequences; | Death |
| | analgesics indicated | prescription analgesics | hospitalization or intervention | symptoms associated with | |
| | | indicated; limiting instrumental | indicated for pain control (e.g., | neurovascular compromise | |
| | | ADL | vertebroplasty); limiting self care | | |
| | | | ADL; disability | | |
| | injury to the spine in which the con | | | | |
| Stenosis of gastrointestinal | - | Symptomatic; IV fluids indicated | Severely altered GI function; | Life-threatening consequences; | Death |
| stoma | | <24 hrs; manual dilation at | tube feeding, TPN or | urgent operative intervention | |
| | | bedside | hospitalization indicated; elective operative intervention | indicated | |
| | | | indicated | | |
| Definition: A finding of parrowing | of the gastrointestinal stoma (surg | l<br>rically created opening on the surf | ı | ļ | 1 |
| Stomal ulcer | Asymptomatic; clinical or | Symptomatic; medical | Severe symptoms; elective | | |
| Storrial dicer | diagnostic observations only; | intervention indicated | operative intervention indicated | - | - |
| | intervention not indicated | intervention interest | operative intervention introduced | | |
| Definition: A disorder characterize | ed by a circumscribed, inflammato | rv and necrotic erosive lesion on t | r<br>he ieiunal mucosal surface close t | o the anastomosis site following a | |
| | , | ., | ···- j-j-·· | | |
| gastroenterostomy procedure. | Minimal blacking at a selficial and | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| 71 | iviinimai bieeding identified on | 1 | indicated; radiologic or | urgent intervention indicated | |
| ,, | Minimal bleeding identified on clinical or diagnostic exam; | intervention indicated | | | 1 |
| ,, | - | intervention indicated | endoscopic intervention | | |
| ,, | clinical or diagnostic exam; | intervention indicated | _ | | |
| Tracheal hemorrhage | clinical or diagnostic exam;<br>intervention not indicated | intervention indicated | endoscopic intervention | | |
| Tracheal hemorrhage Definition: A finding of bleeding from the second control of the se | clinical or diagnostic exam;<br>intervention not indicated | intervention indicated Symptomatic (e.g., noisy airway | endoscopic intervention | Life-threatening airway | Death |
| gastroenterostomy procedure. Tracheal hemorrhage Definition: A finding of bleeding find the struction in the struction is seen that the struction is seen the struction in the struction in the struction is seen the struction in the struction is seen the struction in the struction in the struction in the struction is seen the struction in the struction in the struction is seen the struction in the struction in the struction is seen the struction in the struction in the struction is seen the struction in the struction in the struction is seen the struction in the struction | clinical or diagnostic exam;<br>intervention not indicated | | endoscopic intervention indicated | Life-threatening airway compromise; urgent intervention | Death |
| Tracheal hemorrhage Definition: A finding of bleeding from the second control of the se | clinical or diagnostic exam;<br>intervention not indicated<br>rom the trachea. | Symptomatic (e.g., noisy airway | endoscopic intervention indicated Stridor; radiologic or endoscopic | I | Death |
| Tracheal hemorrhage Definition: A finding of bleeding from the second control of the se | clinical or diagnostic exam; intervention not indicated from the trachea. Partial asymptomatic obstruction on examination | Symptomatic (e.g., noisy airway breathing), no respiratory | endoscopic intervention indicated Stridor; radiologic or endoscopic intervention indicated (e.g., stent, laser); limiting self care | compromise; urgent intervention | Death |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Tracheostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood lea | kage from the tracheostomy site. | | | | |
| Ureteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | lue to breakdown of a ureteral ana | | | | |
| Jrethral anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a urethral ana | stomosis (surgical connection of tw | vo separate anatomic structures). | <u> </u> | |
| Urostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | of contents from a urostomy. | 1 | İ | | |
| Urostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or endoscopic repair or stent placement indicated | Altered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | T. | | | |
| Urostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding | from the urostomy site. | ' | , | • | • |
| Urostomy stenosis | - | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | of the opening of a urostomy. | , | • | • | |
| Uterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a uterine anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a rupture in the uterine wall. | | Cause aumentama, radialagia | Life threatening concessions | Dooth |
| /aginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vaginal anas | stomosis (surgical connection of tw | o separate anatomic structures). | İ | |
| Vas deferens anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vas deferens | s anastomosis (surgical connection | n of two separate anatomic structu | res). | |
| Vascular access complication | - | Device dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including pulmonary embolism or life-threatening thrombus | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Venous injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self care ADL; repair or revision indicated; disabling | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | | I | | I | |
| Wound complication | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound; local care indicated | Hernia without evidence of<br>strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by<br>operative intervention indicated | Hernia with evidence of<br>strangulation; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| Definition: A finding of development | ent of a new problem at the site of | an existing wound. | | | |
| Wound dehiscence | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound with local care; asymptomatic hernia or symptomatic hernia without evidence of strangulation | Fascial disruption or dehiscence without evisceration; primary wound closure or revision by operative intervention indicated | Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| Definition: A finding of separation | of the approximated margins of a | surgical wound. | | | |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of traumatic | injury to the wrist joint in which the | continuity of a wrist bone is broke | en. | | |
| Injury, poisoning and procedural complications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Investigations | <u> </u> | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | | romboplastin time is found to be g | | possible indicator of coagulopat | hy, a prolonged |
| | | s and disorders, both primary and | İ | - 00 0 I II N | |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | | n increase in the level of alanine a | 1 | 1 | |
| Alkaline phosphatase increased | 1 | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | | n increase in the level of alkaline p | · | | 1 |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen. | _ |
| Blood antidiuretic hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of antidiuretic horm | none in the blood specimen. | | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is a | ssociated with jaundice. | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotrop | hin in a blood specimen. | | |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; | Symptomatic; medical intervention indicated; limiting instrumental ADI | Severe symptoms; limiting self care ADL | - | - |
| Definition: A finding based on lab | intervention not indicated | instrumental ADL | armone in a blood enseimen | l | l . |
| | | bnormal levels of gonadotrophin h | ormone in a blood specimen. | | |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of prolactin hormor | ne in a blood specimen. | | • |
| Carbon monoxide diffusing capacity decreased | 3 - 5 units below LLN; for follow-<br>up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | 6 - 8 units below LLN; for follow-<br>up, an asymptomatic decrease<br>of >5 - 8 units (ml/min/mm Hg)<br>below the baseline value | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., >Grade 2 hypoxia or >Grade 2 or higher dyspnea) | - | - |
| Definition: A finding based on lun | g function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | ' | ' |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| | | of cardiac troponin I in a biologica | Ι΄. | I | 1 |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test result | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | | |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | |
| Cholesterol high | | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | oratory test results that indicate h | igher than normal levels of choles | terol in a blood specimen. | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in levels of creatine pho | osphokinase in a blood specimen. | | |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5<br>x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of creatinine in a b | ological specimen. | | |
| Ejection fraction decreased | - | Resting ejection fraction (EF) 50 - 40%; 10 - 19% drop from baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline | Resting ejection fraction (EF) <20% | - |
| Definition: The percentage compo | uted when the amount of blood eje | ected during a ventricular contracti | on of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected interval prolonged | | QTc 481 - 500 ms | QTc >= 501 ms on at least two<br>separate ECGs | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| | | bnormally long corrected QT inter | | | 1 |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75% decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of fibrinogen i | n a blood specimen. | • | • |
| Forced expiratory volume decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on tes | t results that indicate a relative de | crease in the fraction of the forced | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased<br>Definition: A finding based on lab | >ULN - 2.5 x ULN<br>oratory test results that indicate hi | >2.5 - 5.0 x ULN<br>gher than normal levels of the enz | >5.0 - 20.0 x ULN<br>yme gamma-glutamyltransferase | >20.0 x ULN<br>in the blood specimen. GGT (gam | -<br>nma- |
| glutamyltransferase ) catalyzes th | ne transfer of a gamma glutamyl g | roup from a gamma glutamyl pept | de to another peptide, amino acid | s or water. | |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate al | onormal levels of growth hormone | in a biological specimen. | | |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ,<br>n decrease in levels of haptoglobir | in a blood specimen. | • | • |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >2 - 4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | - | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of hemoglobin in a | biological specimen. | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>anticoagulation | >2.5 x ULN; >2.5 times above baseline if on anticoagulation | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the ratio of the patier | t's prothrombin time to a control s | ample in the blood. | |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of lipase in | a biological specimen. | | |
| ymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of lymphocyte | es in a blood specimen. | | |
| ymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormal increase in the numbe | r of lymphocytes in the blood, effu | sions or bone marrow. | |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of neutrophils | in a blood specimen. | | |
| Pancreatic enzymes decreased | <lln and="" asymptomatic<="" td=""><td>Increase in stool frequency,<br/>bulk, or odor; steatorrhea</td><td>Sequelae of absorption deficiency</td><td>-</td><td>-</td></lln> | Increase in stool frequency,<br>bulk, or odor; steatorrhea | Sequelae of absorption deficiency | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of pancreatic | enzymes in a biological specimen. | • | • |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<="" 75,000="" <lln="" mm3;="" td=""><td>&lt;75,000 - 50,000/mm3; &lt;75.0 -</td><td>&lt;50,000 - 25,000/mm3; &lt;50.0 -</td><td>&lt;25,000/mm3; &lt;25.0 x 10e9 /L</td><td>-</td></lln> | <75,000 - 50,000/mm3; <75.0 - | <50,000 - 25,000/mm3; <50.0 - | <25,000/mm3; <25.0 x 10e9 /L | - |
| | 75.0 x 10e9 /L | 50.0 x 10e9 /L | 25.0 x 10e9 /L | | |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the levels of amylase | in a serum specimen. | | |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | - |
| Definition: A finding based on tes | t results that indicate urine produc | tion is less relative to previous ou | tput. | | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value; | <50% of predicted value; | - | - |
| | | limiting instrumental ADL | limiting self care ADL | | |
| Definition: A finding based on pul | monary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | um inhalation) when compared to | the predicted |
| value. | | | | | |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characterized | d by an increase in overall body w | eight; for pediatrics, greater than t | he baseline growth curve. | | |
| Weight loss | 5 to <10% from baseline; | 10 - <20% from baseline; | >=20% from baseline; tube | - | - |
| | intervention not indicated | nutritional support indicated | feeding or TPN indicated | | |
| Definition: A finding characterized | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" td="" x<=""><td>&lt;3000 - 2000/mm3; &lt;3.0 - 2.0 x</td><td>&lt;2000 - 1000/mm3; &lt;2.0 - 1.0 x</td><td>&lt;1000/mm3; &lt;1.0 x 10e9 /L</td><td>-</td></lln> | <3000 - 2000/mm3; <3.0 - 2.0 x | <2000 - 1000/mm3; <2.0 - 1.0 x | <1000/mm3; <1.0 x 10e9 /L | - |
| | 10e9 /L | 10e9 /L | 10e9 /L | | |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in number of white blo | od cells in a blood specimen. | · | |
| Investigations - Other, specify | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| | , , , | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated;<br>disabling; limiting self care ADL | | |
| | | 1 | uisabiing, iiiniiing seil cale ADL | l . | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| cidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| efinition: A disorder characteri | zed by abnormally high acidity (high | h hydrogen-ion concentration) of t | he blood and other body tissues. | Т | |
| Alcohol intolerance | - | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an increase in sensitivity to | the adverse effects of alcohol, wh | ich can include nasal congestion, | skin flushes, heart dysrhythmias, i | nausea, |
| omiting, indigestion and heada<br>Alkalosis | pH >normal, but <=7.5 | | pH >7.5 | Life threatening consequences | Death |
| | | -<br> | 1. | Life-threatening consequences | Deam |
| | zed by abnormally high alkalinity (k | | | | D#- |
| Anorexia | Loss of appetite without alteration in eating habits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a loss of appetite. | | | | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by excessive loss of water from | n the body. It is usually caused by | severe diarrhea, vomiting or diaph | noresis. | |
| Glucose intolerance | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an inability to properly meta | bolize glucose. | | | |
| Hypercalcemia | Corrected serum calcium of<br>>ULN - 11.5 mg/dL; >ULN - 2.9<br>mmol/L; Ionized calcium >ULN<br>- 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of calcium (corrected for all | oumin) in blood. | |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteri<br>ntolerance. | zed by laboratory test results that in | ndicate an elevation in the concen | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucose |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri<br>he use of diuretic drugs. | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of potassium in the blood; a | associated with kidney failure or so | ometimes w |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23<br>mmol/L | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate an elevation in the concen | tration of magnesium in the blood | · | 1 |
| lypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| | zed by laboratory test results that in | | | T | 1 |
| ypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4 mmol/L;<br>life-threatening consequences | Death |
| | zed by laboratory test results that in | ndicate an elevation in the concen | 1 | | 1 |
| yperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| efinition: A disorder characteri | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of uric acid. | | |
| ypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteri | ्।<br>zed by laboratory test results that ir | ndicate a low concentration of albu | umin in the blood. | • | • |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -="" 1.0="" l<="" mmol="" td=""><td>Corrected serum calcium of<br/>&lt;8.0 - 7.0 mg/dL; &lt;2.0 - 1.75<br/>mmol/L; lonized calcium &lt;1.0 -<br/>0.9 mmol/L; symptomatic</td><td>Corrected serum calcium of &lt;7.0 - 6.0 mg/dL; &lt;1.75 - 1.5 mmol/L; lonized calcium &lt;0.9 - 0.8 mmol/L; hospitalization indicated</td><td>Corrected serum calcium of<br/>&lt;6.0 mg/dL; &lt;1.5 mmol/L;<br/>lonized calcium &lt;0.8 mmol/L;<br/>life-threatening consequences</td><td>Death</td></lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 - 6.0 mg/dL; <1.75 - 1.5 mmol/L; lonized calcium <0.9 - 0.8 mmol/L; hospitalization indicated | Corrected serum calcium of<br><6.0 mg/dL; <1.5 mmol/L;<br>lonized calcium <0.8 mmol/L;<br>life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate a low concentration of calc | ium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0<br="" 55="" <lln="" dl;="" mg="">mmol/L</lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of gluc | ose in the blood. | | |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate a low concentration of pota | assium in the blood. | | |
| Hypomagnesemia | <lln -="" 0.5="" 1.2="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3 mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3 mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of mag | nesium in the blood. | | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate a low concentration of sod | um in the blood. | | |
| Hypophosphatemia | <lln -="" 0.8<br="" 2.5="" <lln="" dl;="" mg="">mmol/L</lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6 mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3 mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate a low concentration of pho | sphates in the blood. | | |
| Iron overload | - | Moderate symptoms; intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by accumulation of iron in the t | issues. | | | |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| Definition: A disorder characteriz | ed by having a high amount of boo | dy fat. | | | |
| Tumor lysis syndrome | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by metabolic abnormalities that | t result from a spontaneous or the | rapy-related cytolysis of tumor cell | S | |
| Metabolism and nutrition disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the abdomir | nal wall. | | |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in a joint. | T | T | |
| Arthritis | Mild pain with inflammation, erythema, or joint swelling | Moderate pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inflammation involving a joir | nt. | i | i | |
| Avascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by necrotic changes in the bond<br>d the destruction of the bone struc | | od supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the back region. | | | |
| Bone pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the bones. | 1 | | |
| Buttock pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the buttocks. | | | |
| Chest wall pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the chest wall region. | | T | |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth o | of bone. | | • | |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the | deep connective tissues. | 1 | | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n on the lateral side of the body in | the region below the ribs and abo | ve the hip. | |
| Generalized muscle weakness | Symptomatic; weakness<br>perceived by patient but not<br>evident on physical exam | Symptomatic; weakness evident on physical exam; weakness limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | - |
| | ed by a reduction in the strength o | | | | |
| Growth suppression | Reduction in growth velocity by 10 - 29% ideally measured over the period of a year ed by of stature that is smaller that | Reduction in growth velocity by 30 - 49% ideally measured over the period of a year or 0 - 49% reduction in growth from the baseline growth curve | Reduction in growth velocity of >=50% ideally measured over the period of a year | - | - |

| Musculoskeletal and connective tissue disorders Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Head soft tissue necrosis | | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the head. | | | |
| Joint effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated; disabling | - | - |
| Definition: A disorder characteriz | ed by excessive fluid in a joint, usu | ually as a result of joint inflammati | on. | I | |
| Joint range of motion decreased | <=25% loss of ROM (range of<br>motion); decreased ROM<br>limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50% decrease in ROM; limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a decrease in joint flexibility | of any joint. | | | |
| Joint range of motion decreased cervical spine | Mild restriction of rotation or flexion between 60 - 70 degrees | Rotation <60 degrees to right or left; <60 degrees of flexion | Ankylosed/fused over multiple segments with no C-spine rotation | - | - |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | cervical spine joint. | ī | ř | |
| Joint range of motion decreased lumbar spine | Stiffness; difficulty bending to the floor to pick up a very light object but able to do athletic activity | Pain with range of motion<br>(ROM) in lumbar spine; requires<br>a reaching aid to pick up a very<br>light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>ankylosis or fused over multiple<br>segments with no L-spine<br>flexion (e.g., unable to reach to<br>floor to pick up a very light<br>object) | - | - |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | lumbar spine joint. | | | |
| Kyphosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the thoracic portion of | of the spine. | | |
| Lordosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the lumbar portion of | the spine. | | |
| Muscle weakness left-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the left side of th | e body. | | |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the lower limb muscles. | | | |
| Muscle weakness right-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the right side of | the body. | | 1 |
| Muscle weakness trunk | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| | | • | • | • | • |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the trunk muscles. | | | |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g.,<br>shoe insert) or covered by<br>clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; disabling | - | - |
| Definition: A disorder characteri | zed by of a malformation of the mu | sculoskeletal system. | ļ | ! | • |
| Myalgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | | |
| Myositis | Mild pain | Moderate pain associated with weakness; pain limiting instrumental ADL | Pain associated with severe weakness; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by inflammation involving the s | keletal muscles. | | | |
| Neck pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the neck area. | 1 | T | |
| Neck soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the soft tissues of the neck. | | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of osteoporosis or Bone Mineral Density (BMD) t-score -1 to -2.5 (osteopenia); no loss of height or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm;<br>hospitalization indicated; limiting<br>self care ADL | - | - |
| Definition: A disorder characteri composition), resulting in increa | ized by reduced bone mass, with a ased fracture incidence. | decrease in cortical thickness and | I in the number and size of the trab | peculae of cancellous bone (but no | rmal chen |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the upper or lower extremities | S | | |
| Pelvic soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a necrotic process occurring | | 1 | | |
| Scoliosis | <20 degrees; clinically undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | - | - |
| Definition: A disorder characteri | zed by a malformed, lateral curvatu | re of the spine. | 1 | 1 | |
| Soft tissue necrosis lower limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the soft tissues of the lower ex | tremity. | | |
| Soft tissue necrosis upper limb | - | Local wound care; medical intervention indicated (e.g., dressings or topical | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap | Life-threatening consequences; urgent intervention indicated | Death |

| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to slide skin, unable to pinch skin; limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characterize | ed by fibrotic degeneration of the s | superficial soft tissues. | | | _ |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, soft foods or purees | Decreased ROM with inability to adequately aliment or hydrate orally | - | - |
| Definition: A disorder characterize | ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | mastication. | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - 5 cm; shoe lift indicated; limiting instrumental ADL | | - | - |
| Definition: A disorder characterize | ed by of a discrepancy between th | e lengths of the lower or upper ex | tremities. | | |
| Musculoskeletal and connective tissue disorder - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Neoplasms benig | n, malignant and unspec | cified (incl cysts and poly | yps) | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Leukemia secondary to oncology chemotherapy | - | - | - | Present | Death |
| Definition: A disorder characterize | ed by leukemia arising as a result | of the mutagenic effect of chemot | herapy agents. | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by insufficiently healthy hemata | poietic cell production by the bone | e marrow. | | |
| Treatment related secondary malignancy | - | - | Non life-threatening secondary malignancy | Acute life-threatening secondary malignancy; blast crisis in leukemia | Death |
| Definition: A disorder characterize | ed by development of a malignanc | by most probably as a result of trea | atment for a previously existing ma | alignancy. | |
| Tumor pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort from a ne | eoplasm that may be pressing on | a nerve, blocking blood vessels, ir | nflamed or fractured from metastas | sis. |
| Neoplasms benign, malignant<br>and unspecified (incl cysts and<br>polyps) - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Adverse Event Abducens nerve disorder Definition: A disorder characterize Accessory nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | 2 Moderate symptoms; limiting | Grade 3 | 4 | 5 |
|---|---|---|---|---|---|
| Abducens nerve disorder<br>Definition: A disorder characterize | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | | 3 | 4 | 5 |
| Definition: A disorder characterize | diagnostic observations only; intervention not indicated | Moderate symptoms; limiting | | | , |
| | | instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Accessory nerve disorder | ed by involvement of the abducens | s nerve (sixth cranial nerve). | I | | |
| | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by involvement of the accessor | y nerve (eleventh cranial nerve). | | | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by involvement of the acoustic | nerve (eighth cranial nerve). | | | |
| Akathisia | Mild restlessness or increased motor activity | Moderate restlessness or increased motor activity; limiting instrumental ADL | Severe restlessness or increased motor activity; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an uncomfortable feeling of | inner restlessness and inability to | stay still; this is a side effect of sor | me psychotropic drugs. | |
| Amnesia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss;<br>limiting self care ADL | - | - |
| | ed by systematic and extensive lo | ss of memory. | <u> </u> | | |
| Aphonia | - | - | Voicelessness; unable to speak | - | - |
| | ed by the inability to speak. It may | | | | l |
| Arachnoiditis | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by inflammation of the arachno | , | 1 | | |
| Ataxia | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | - | - |
| Definition: A disorder characterize | ed by lack of coordination of musc | le movements resulting in the imp | airment or inability to perform volu | ntary activities. | |
| Brachial plexopathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by regional paresthesia of the b | orachial plexus, marked discomfor | t and muscle weakness, and limite | ed movement in the arm or hand. | |
| Central nervous system necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; corticosteroids indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a necrotic process occurring | in the brain and/or spinal cord. | | <u> </u> | |
| Cerebrospinal fluid leakage | Post-craniotomy: asymptomatic;<br>Post-lumbar puncture: transient<br>headache; postural care<br>indicated | Post-craniotomy: moderate<br>symptoms; medical intervention<br>indicated; Post-lumbar<br>puncture: persistent moderate<br>symptoms; blood patch<br>indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by loss of cerebrospinal fluid in | to the surrounding tissues. | T | <b>I</b> | |
| Cognitive disturbance | Mild cognitive disability; not<br>interfering with work/school/life<br>performance; specialized<br>educational services/devices<br>not indicated | Moderate cognitive disability;<br>interfering with work/school/life<br>performance but capable of<br>independent living; specialized<br>resources on part time basis<br>indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | - | - |
| Definition: A disorder characterize | ed by a conspicuous change in co | gnitive function. | T . | <u> </u> | 1 |
| Concentration impairment | Mild inattention or decreased level of concentration | Moderate impairment in attention or decreased level of concentration; limiting instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | - | - |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to stimuli; limiting instrumental ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ा<br>zed by a decrease in ability to perc | | I | l | I |
| Dizziness | Mild unsteadiness or sensation of movement | Moderate unsteadiness or sensation of movement; limiting instrumental ADL | Severe unsteadiness or sensation of movement; limiting self care ADL | - | - |
| Definition: A disorder characterize | '<br>zed by a disturbing sensation of lig | htheadedness, unsteadiness, gidd | liness, spinning or rocking. | ' | |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characterization | zed by slow and slurred speech res | sulting from an inability to coordina | ate the muscles used in speech. | I | 1 |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation. | Г | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet<br>(e.g., oral supplements);<br>noxious or unpleasant taste;<br>loss of taste | - | - | - |
| Definition: A disorder characteriz | zed by abnormal sensual experien | ce with the taste of foodstuffs; it ca | n be related to a decrease in the s | sense of smell. | |
| Dysphasia | Awareness of receptive or expressive characteristics; not impairing ability to communicate | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | - | - |
| Definition: A disorder characterize | zed by impairment of verbal comm | unication skills, often resulting fron | n brain damage. | T | 1 |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | - |
| Definition: A disorder characterize | zed by swelling due to an excessiv | e accumulation of fluid in the brain | l.<br>T | T | 1 |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a pathologic process involvi | | | l . | 1 |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary movements; limiting instrumental ADL | Severe involuntary movements or torticollis; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by abnormal, repetitive, involu | ntary muscle movements, frenzied | speech and extreme restlessness | ·<br>i. | |
| Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterization | zed by a reduction in the strength o | of the facial muscles. | | T | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the facial ne | rve (seventh cranial nerve). | 1 | | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by involvement of the glossoph | naryngeal nerve (ninth cranial nerv | e). | | |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | omfort in various parts of the head | , not confined to the area of distrib | ution of any nerve. | 1 |
| Hydrocephalus | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; intervention not indicated | Severe symptoms or neurological deficit; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal increase of ce | rebrospinal fluid in the ventricles o | f the brain. | | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for | Severe increased need for | - | - |

| | 1 | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the hypoglos | sal nerve (twelfth cranial nerve). | , | | • |
| Intracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the cranium. | | | | |
| schemia cerebrovascular | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | - | - | - |
| Definition: A disorder characteriz<br>damage. | red by a decrease or absence of bl | ood supply to the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | ological |
| Vth nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the trochlear | nerve (fourth cranial nerve). | 1 | 1 | |
| Lethargy | Mild symptoms; reduced alertness and awareness | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A disorder characteriz | zed by a decrease in consciousnes | s characterized by mental and phy | ysical inertness. | T | |
| Leukoencephalopathy | Asymptomatic; small focal T2/FLAIR hyperintensities; involving periventricular white matter or <1/3 of susceptible areas of cerebrum +/- mild increase in subarachnoid space (SAS) and/or mild ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/3 to 2/3 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate ventriculomegaly | +/- moderate to severe increase | Life-threatening consequences; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Death |
| Definition: A disorder characteriz | ed by diffuse reactive astrocytosis | with multiple areas of necrotic foo | i without inflammation. | | |
| Memory impairment | Mild memory impairment | Moderate memory impairment; limiting instrumental ADL | Severe memory impairment;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by a deterioration in memory fu | inction. | | | |
| Meningismus | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by neck stiffness, headache, ar | nd photophobia resulting from irrit | ation of the cerebral meninges. | | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | red by uncontrolled and purposeles | ss movements. | | 1 | |
| Myelitis | Asymptomatic; mild signs (e.g.,<br>Babinski's reflex or Lhermitte's<br>sign) | Moderate weakness or sensory loss; limiting instrumental ADL | Severe weakness or sensory loss; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by inflammation involving the s | | | marked discomfort and incontined | nce. |
| Neuralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | red by intense painful sensation ald | | I | I | |
| Nystagmus | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involuntary movements of th | ne eyeballs.<br>T | T | T | 1 |
| Oculomotor nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the oculomor | tor nerve (third cranial nerve). | | | |
| Olfactory nerve disorder | - | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize are experienced in the absence of | • | ensory neurons resulting in abnorr | nal cutaneous sensations of tinglir | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation or degeneration | n of the peripheral motor nerves. | | | |
| Peripheral sensory neuropathy | Asymptomatic; loss of deep tendon reflexes or paresthesia | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation or degeneratio | n of the peripheral sensory nerves | S.<br>T | | |
| Phantom pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort related to | o a limb or an organ that is remove | ed from or is not physically part of | the body. | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| Definition: A disorder characterize | ed by an episode of lightheadedne | ess and dizziness which may prece | ede an episode of syncope. | | |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by dysfunction of the corticospi<br>nd a decrease in fine motor coord | | cord. Symptoms include an incre | ease in the muscle tone in the lower | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting instrumental ADL; medical intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize connecting nerve root. | ed by inflammation involving a ner | ve root. Patients experience mark | ed discomfort radiating along a ne | rve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by paralysis of the recurrent lar | yngeal nerve. | | | |
| Reversible posterior leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very<br>abnormal imaging studies;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | | = | | indings of posterior leukoencephal<br>s an acute or subacute reversible o | |
| Seizure | Brief partial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characterize | ed by a sudden, involuntary skelet | tal muscular contractions of cerebr | al or brain stem origin. | | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort in the fac | ce, between the eyes, or upper tee | th originating from the sinuses. | | |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by characterized by excessive | sleepiness and drowsiness. | | | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle tone and increase in resistance through range of motion | Severe increase in muscle tone and increase in resistance through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characterize disturbances. | ed by increased involuntary muscl | e tone that affects the regions inte | ' | It results in gait, movement, and s | peech |
| Stroke | Asymptomatic or mild neurologic deficit; radiographic findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a sudden loss of sensory fu | nction due to an intracranial vascu | lar event. | i . | |
| Syncope Definition: A disorder characterize | d by spontaneous loss of consoir | - | Fainting; orthostatic collapse | - | - |
| Deminition. A disorder characterize | eu by sportaneous loss of consci | ousness caused by insufficient blo | ou supply to the blatt. | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with or without imaging confirmation | - | - | - |
| Definition: A disorder characteriz | ed by a brief attack (less than 24 h | nours) of cerebral dysfunction of va | ascular origin, with no persistent n | eurological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by the uncontrolled shaking mo | ovement of the whole body or indiv | ridual parts. | | |
| Trigeminal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the trigemina | al nerve (fifth cranial nerve). | | | |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the vagus ne | erve (tenth cranial nerve). | • | • | |
| Vasovagal reaction | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz increase in the stimulation of the | ed by a sudden drop of the blood progression vagus nerve. | pressure, bradycardia, and periph | eral vasodilation that may lead to l | oss of consciousness. It results fro | om an |
| Nervous system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Pregna | ancy, puerperium and pe | rinatal conditions | | |
|---|---|---|---|---|
| | | Grade | | |
| 1 | 2 | 3 | 4 | 5 |
| - | - | - | - | Fetal loss at<br>any<br>gestational<br>age |
| ed by death in utero; failure of the | product of conception to show evi | dence of respiration, heartbeat, or | definite movement of a voluntary | muscle after |
| t possibility of resuscitation. | | | | |
| - | <10% percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | - |
| ed by inhibition of fetal growth resu | ulting in the inability of the fetus to | achieve its potential weight. | | |
| , | Delivery of a liveborn infant at >28 to 34 weeks gestation | Delivery of a liveborn infant at 24 to 28 weeks gestation | Delivery of a liveborn infant at 24 weeks of gestation or less | - |
| ed by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | tween the twentieth and thirty-sev | enth week of |
| - | - | Unintended pregnancy | - | - |
| ed by an unexpected pregnancy at | t the time of conception. | ! | ! | ' |
| symptoms; clinical or diagnostic | | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | ted by death in utero; failure of the expossibility of resuscitation. - ted by inhibition of fetal growth resurce of the expossibility of resuscitation. - ted by inhibition of fetal growth resurce of the exposure of a liveborn infant at seven the exposure of a viable infant be exposed by an unexpected pregnancy at the exposure of | ted by death in utero; failure of the product of conception to show evice possibility of resuscitation. - | to d by death in utero; failure of the product of conception to show evidence of respiration, heartbeat, or at possibility of resuscitation. - <10% percentile of weight for gestational age <5% percentile of weight for gestational age <a href="#sectional age">death by inhibition of fetal growth resulting in the inability of the fetus to achieve its potential weight.</a> Delivery of a liveborn infant at Delivery of a liveborn infant at >28 to 34 weeks gestation >28 to 34 weeks gestation >24 to 28 weeks gestation >24 to 28 weeks gestation >25 to 34 weeks gestation >26 to 34 weeks gestation >27 to 34 to 37 weeks gestation >28 to 34 weeks gestation >28 to 34 weeks gestation >28 to 34 weeks gestation >29 to 34 weeks gestation >29 to 34 weeks gestation >29 to 34 weeks gestation >20 to 34 weeks gestat | The destance of the product of conception to show evidence of respiration, heartbeat, or definite movement of a voluntary possibility of resuscitation. - <10% percentile of weight for gestational age <5% percentile of weight for gestational age <1% perc |

| | | Psychiatric disor | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation; hospitalization not indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by a state of restlessness asso | | irritability and tension. | | |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by an inability to achieve orgas | | | | |
| Anxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization not indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder characte stimulus. | erized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dys | pnea unattached to a clearly ident | tifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by a lack of clear and orderly the | nought and behavior. | | | |
| Delayed orgasm | Delay in achieving orgasm not adversely affecting relationship | Delay in achieving orgasm adversely affecting relationship | - | - | - |
| | erized by sexual dysfunction characte | | <u> </u> | I | I_ |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder character reversible condition. | erized by the acute and sudden devel | opment of confusion, illusions, mo | ovement changes, inattentiveness, | agitation, and hallucinations. Usu | ally, it is a |
| Delusions | - | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by false personal beliefs held o | ontrary to reality, despite contradi | ctory evidence and common sense | e. | |
| Depression | Mild depressive symptoms | Moderate depressive symptoms; limiting instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by melancholic feelings of grief | or unhappiness. | , | | , |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | - |
| Definition: A disorder characte | erized by an exaggerated feeling of w | ell-being which is disproportionate | to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by a false sensory perception i | n the absence of an external stimu | ılus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling<br>asleep, staying asleep or<br>waking up early | - | - |
| Definition: A disorder characte | erized by difficulty in falling asleep and | d/or remaining asleep. | 1 | 1 | |
| Libido decreased | Decrease in sexual interest not adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by a decrease in sexual desire | T | T | T | |
| Libido increased | Mild increase in sexual interest<br>not adversely affecting<br>relationship | Moderate increase in sexual interest adversely affecting relationship | Severe increase in sexual interest leading to dangerous behavior | - | - |
| Definition: A disorder characte | erized by an increase in sexual desire | ). | | | |
| Mania | Mild manic symptoms (e.g.,<br>elevated mood, rapid thoughts,<br>rapid speech, decreased need<br>for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by excitement of psychotic pro | portions manifested by mental and | d physical hyperactivity, disorganiz | ation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |

| | | Psychiatric disord | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by a conspicuous change in a p | person's behavior and thinking. | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characterize tumor. | ed by personality change, impaired | d functioning, and loss of touch wi | th reality. It may be a manifestatio | n of schizophrenia, bipolar disord | er or brain |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an inability to rest, relax or b | e still. | | | |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide<br>with serious intent to die which<br>requires hospitalization | - |
| Definition: A disorder characterize | ed by thoughts of taking one's owr | n life. | | | |
| Suicide attempt | - | - | Suicide attempt or gesture without intent to die which may not require hospitalization | Suicide attempt with intent to die which requires hospitalization | Death |
| Definition: A disorder characterize | ed by self-inflicted harm in an atter | mpt to end one's own life. | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |

| Definition: A disorder characterized causes (ureteral or bladder outflow Bladder perforation Definition: A disorder characterized Bladder spasm Definition: A disorder characterized Chronic kidney disease | w obstruction). d by a rupture in the bladder wall. | baseline | Intraperitoneal perforation; | 4 Life-threatening consequences; dialysis indicated ney), renal (kidney damage) and p | 5<br>Death |
|---|---|---|---|---|---|
| Acute kidney injury Definition: A disorder characterized causes (ureteral or bladder outflow Bladder perforation Definition: A disorder characterized Bladder spasm Definition: A disorder characterized Chronic kidney disease | Creatinine level increase of >0.3 mg/dL; creatinine 1.5 - 2.0 x above baseline d by the acute loss of renal function obstruction). | Creatinine 2 - 3 x above baseline on and is traditionally classified as Extraperitoneal perforation, | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated s pre-renal (low blood flow into kid Intraperitoneal perforation; | Life-threatening consequences; dialysis indicated | Death |
| Definition: A disorder characterized causes (ureteral or bladder outflow Bladder perforation Definition: A disorder characterized Bladder spasm Definition: A disorder characterized Chronic kidney disease | mg/dL; creatinine 1.5 - 2.0 x above baseline d by the acute loss of renal functi w obstruction) d by a rupture in the bladder wall. | baseline on and is traditionally classified as Extraperitoneal perforation, | mg/dL; hospitalization indicated s pre-renal (low blood flow into kid | dialysis indicated | |
| causes (ureteral or bladder outflow Bladder perforation Definition: A disorder characterizer Bladder spasm Definition: A disorder characterizer Chronic kidney disease | w obstruction). d by a rupture in the bladder wall. | Extraperitoneal perforation, | Intraperitoneal perforation; | I | |
| Definition: A disorder characterizer Bladder spasm Definition: A disorder characterizer Chronic kidney disease | | | · · | | |
| Bladder spasm Definition: A disorder characterized Chronic kidney disease | | | elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder characterized | | | | <u> </u> | 1 |
| Chronic kidney disease | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | - | - |
| * | d by a sudden and involuntary co | ntraction of the bladder wall. | | | |
| 1 | eGFR (estimated Glomerular<br>Filtration Rate) or CrCl<br>(creatinine clearance) <lln -="" 60<br="">ml/min/1.73 m2 or proteinuria<br/>2+ present; urine<br/>protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated | Death |
| Definition: A disorder characterized | d by gradual and usually permane | ent loss of kidney function resulting | ng in renal failure. | | 1 |
| i | Microscopic hematuria; minimal increase in frequency, urgency, dysuria, or nocturia; new onset of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder characterized | d by inflammation of the bladder | which is not caused by an infectio | n of the urinary tract. | • | • |
| | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characterized | d by laboratory test results that in | dicate blood in the urine. | | <b>.</b> | |
| | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characterize | d by laboratory test results that in | dicate the presence of free hemo | globin in the urine. | | |
| | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 - 3.4 g/24 hrs;<br>Pediatric: urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5<br>g/24 hrs;<br>Pediatric: urine P/C >1.9 | - | - |
| Definition: A disorder characterize | d by laboratory test results that in | dicate the presence of excessive | protein in the urine. It is predomina | antly albumin, but also globulin. | |
| \$ | Asymptomatic or mild symptoms; occasional use of nonprescription analgesics indicated | Symptomatic; oral antiemetics indicated; around the clock nonprescription analgesics or any oral narcotic analgesics indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences;<br>urgent radiologic, endoscopic or<br>operative intervention indicated | Death |
| Definition: A disorder characterized | d by the formation of crystals in the | ne pelvis of the kidney. | T | Γ | |
| 1 | Mild pain not interfering with<br>activity; nonprescription<br>medication indicated | Moderate pain; limiting instrumental ADL; prescription medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |

| | | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or hospitalization indicated; elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the kidney. | | | | |
| Urinary fistula | - | Noninvasive intervention indicated; urinary or suprapubic catheter placement indicated | Limiting self care ADL; elective radiologic, endoscopic or operative intervention indicated; permanent urinary diversion indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | ized by an abnormal communication | between any part of the urinary s | system and another organ or anato | omic site. | |
| Urinary frequency | Present | Limiting instrumental ADL; medical management indicated | - | - | - |
| Definition: A disorder character | rized by urination at short intervals. | T | T | T | т |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g.,<br>clamp, collagen injections);<br>operative intervention indicated;<br>limiting self care ADL | - | - |
| Definition: A disorder character | ized by inability to control the flow o | f urine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder character | ized by accumulation of urine within | the bladder because of the inabil | ity to urinate. | • | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of contents of the urinary tract. | 1 | T | |
| Urinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by a sensation of marked disco | omfort in the urinary tract. | 1 | 1 | |
| Urinary urgency | Present | Limiting instrumental ADL;<br>medical management indicated | - | - | - |
| Definition: A disorder character | ized by a sudden compelling urge to | o urinate. | 1 | | |
| Urine discoloration | Present | - | - | - | - |
| Definition: A disorder character | ized by a change in the color of the | urine. | | | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Rep | productive system and bi | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azoospermia | - | - | Absence of sperm in ejaculate | - | - |
| Definition: A disorder character | rized by laboratory test results that in | ndicate complete absence of sperr | matozoa in the semen. | | |
| Breast atrophy | Minimal asymmetry; minimal | Moderate asymmetry; moderate | Asymmetry >1/3 of breast | - | - |
| | atrophy | atrophy | volume; severe atrophy | | |
| Definition: A disorder character | rized by underdevelopment of the bre | east. | | • | |
| Breast pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder character | rized by marked discomfort sensation | n in the breast region. | , | • | |
| Dysmenorrhea | Mild symptoms; intervention not | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| , | indicated | instrumental ADL | care ADL | | |
| Definition: A disorder character | rized by abnormally painful abdomina | al cramps during menses. | ! | ! | |
| Dyspareunia | Mild discomfort or pain | Moderate discomfort or pain | Severe discomfort or pain | _ | I _ |
| 3 y o paro a ma | associated with vaginal | associated with vaginal | associated with vaginal | | |
| | penetration; discomfort relieved | penetration; discomfort or pain | penetration; discomfort or pain | | |
| | with use of vaginal lubricants or | partially relieved with use of | unrelieved by vaginal lubricants | | |
| | estrogen | vaginal lubricants or estrogen | or estrogen | | [ |
| Definition: A disorder character | rized by painful or difficult coitus. | | | | |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde | - | - | - |
| | | ejaculation | | | |
| Definition: A disorder character | rized by problems related to ejaculati | ion. This category includes prema | ture, delayed, retrograde and pain | ful ejaculation. | |
| Erectile dysfunction | Decrease in erectile function | Decrease in erectile function | Decrease in erectile function | = | - |
| , | (frequency or rigidity of | (frequency/rigidity of erections), | (frequency/rigidity of erections) | | |
| | erections) but intervention not | erectile intervention indicated, | but erectile intervention not | | |
| | indicated (e.g., medication or | (e.g., medication or mechanical | helpful (e.g., medication or | | |
| | use of mechanical device, | devices such as penile pump) | mechanical devices such as | | |
| | penile pump) | | penile pump); placement of a | | |
| | | | permanent penile prosthesis | | |
| | | | indicated (not previously present) | | |
| Definition: A disorder character | ।<br>rized by the persistent or recurrent in | l<br>pability to achieve or to maintain a | | l | ı |
| Fallopian tube obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder character | rized by blockage of the normal flow | ı | 1 - | | I |
| Delimition. A disorder character | | or the contents in the falloplan tur. | | | |
| | 1 | 0 1 2 12 1 2 | | | |
| Fallopian tube stenosis | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| Fallopian tube stenosis | Asymptomatic clinical or diagnostic observations only; | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | urgent operative intervention | Death |
| · | Asymptomatic clinical or diagnostic observations only; intervention not indicated | not indicated | | I | Death |
| | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian | not indicated | operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) | |
| · | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian saymptomatic clinical or | not indicated tube lumen. Symptomatic and intervention | operative intervention indicated Severe symptoms; elective | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; | Death |
| Definition: A disorder characte | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian symptomatic clinical or diagnostic observations only; | not indicated | operative intervention indicated Severe symptoms; elective | urgent operative intervention indicated (e.g., organ resection) | |
| Definition: A disorder character<br>Female genital tract fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian Asymptomatic clinical or diagnostic observations only; intervention not indicated | not indicated tube lumen. Symptomatic and intervention not indicated | operative intervention indicated Severe symptoms; elective operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by an abnormal communication | tube lumen. Symptomatic and intervention not indicated | operative intervention indicated Severe symptoms; elective operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical | operative intervention indicated Severe symptoms; elective operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of th | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated | Severe symptoms; elective operative intervention indicated system organ and another organ or - | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of secondarians. | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated ary female sex characteristics in m | Severe symptoms; elective operative intervention indicated very stem organ and another organ or an ales due to extrinsic factors. | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of of secondarized Mild swelling or obscuration of | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated ary female sex characteristics in m Readily apparent obscuration of | Severe symptoms; elective operative intervention indicated vystem organ and another organ or alles due to extrinsic factors. | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of secondarized mild swelling or obscuration of anatomic architecture on close | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated ary female sex characteristics in m Readily apparent obscuration of anatomic architecture; | Severe symptoms; elective operative intervention indicated vystem organ and another organ or each state of the system organ and another organ or each state of the system organ and another organ or each state of the system organ and another organ or each system organ and each state of the system or each sy | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of of secondarized Mild swelling or obscuration of | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated ary female sex characteristics in m Readily apparent obscuration of anatomic architecture; obliteration of skin folds; readily | Severe symptoms; elective operative intervention indicated vystem organ and another organ or alles due to extrinsic factors. | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of secondarized mild swelling or obscuration of anatomic architecture on close | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated ary female sex characteristics in m Readily apparent obscuration of anatomic architecture; obliteration of skin folds; readily apparent deviation from normal | Severe symptoms; elective operative intervention indicated vystem organ and another organ or each state of the system organ and another organ or each state of the system organ and another organ or each state of the system organ and another organ or each system organ and each state of the system or each sy | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of anatomic architecture on close inspection | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive s Moderate symptoms; medical intervention indicated ary female sex characteristics in m Readily apparent obscuration of anatomic architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour | Severe symptoms; elective operative intervention indicated system organ and another organ or elective operative intervention indicated system organ and another organ or election organ and election organ organization from normal anatomic contour; limiting self care ADL | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of secondarized mild swelling or obscuration of anatomic architecture on close inspection | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive symptoms; medical intervention indicated ary female sex characteristics in machine architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour accumulation of fluid in the genit | Severe symptoms; elective operative intervention indicated severe symptoms; elective operative intervention indicated system organ and another organ or electrons. Lymphorrhea; gross deviation from normal anatomic contour; limiting self care ADL | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by swelling or obscuration of anatomic architecture on close inspection | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive symptoms; medical intervention indicated ary female sex characteristics in machine architecture; obliteration of shin folds; readily apparent deviation from normal anatomic contour accumulation of fluid in the genite symptomatic (e.g., pain or | Severe symptoms; elective operative intervention indicated operati | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema Definition: A disorder character Genital edema | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by swelling or obscuration of anatomic architecture on close inspection | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive semantic | Severe symptoms; elective operative intervention indicated severe symptoms; elective operative intervention indicated system organ and another organ or electrons. Lymphorrhea; gross deviation from normal anatomic contour; limiting self care ADL | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema Definition: A disorder character Gynecomastia Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of th | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive symptoms; medical intervention indicated ary female sex characteristics in manatomic architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour accumulation of fluid in the genit symptomatic (e.g., pain or psychosocial impact) ne breasts in males. | Severe symptoms; elective operative intervention indicated system organ and another organ or all ales due to extrinsic factors. Lymphorrhea; gross deviation from normal anatomic contour; limiting self care ADL als. Severe symptoms; elective operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated anatomic site. | Death - |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema Definition: A disorder character Gynecomastia Definition: A disorder character | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of diagnostic observations only; intervention not indicated rized by an abnormal communication Mild symptoms; intervention not indicated rized by the development of secondarized by the development of secondarized by the development of secondarized by the development of secondarized by swelling or obscuration of anatomic architecture on close inspection | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive semantic | Severe symptoms; elective operative intervention indicated system organ and another organ or alles due to extrinsic factors. Lymphorrhea; gross deviation from normal anatomic contour; limiting self care ADL Severe symptoms; elective operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated anatomic site. - Life-threatening consequences; | |
| Definition: A disorder character Female genital tract fistula Definition: A disorder character Feminization acquired Definition: A disorder character Genital edema Definition: A disorder character Genital edema | Asymptomatic clinical or diagnostic observations only; intervention not indicated rized by a narrowing of the fallopian of th | not indicated tube lumen. Symptomatic and intervention not indicated between a female reproductive symptoms; medical intervention indicated ary female sex characteristics in manatomic architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour accumulation of fluid in the genit symptomatic (e.g., pain or psychosocial impact) ne breasts in males. | Severe symptoms; elective operative intervention indicated system organ and another organ or all ales due to extrinsic factors. Lymphorrhea; gross deviation from normal anatomic contour; limiting self care ADL als. Severe symptoms; elective operative intervention indicated | urgent operative intervention indicated (e.g., organ resection) Life-threatening consequences; urgent intervention indicated anatomic site. | Death - |

| | Rep | productive system and bi | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | red by the presence of blood in a fa | | <u> </u> | | 1 |
| Irregular menstruation | Intermittent menses with skipped menses for no more than 1 to 3 months | Intermittent menses with skipped menses for more than 4 to 6 months | Persistent amenorrhea for more than 6 months | - | - |
| Definition: A disorder characteriz | ed by irregular cycle or duration of | | T | | |
| Lactation disorder | Mild changes in lactation, not significantly affecting production or expression of breast milk | Changes in lactation,<br>significantly affecting breast<br>production or expression of<br>breast milk | - | - | - |
| Definition: A disorder characteriz | ed by disturbances of milk secretion | on. It is not necessarily related to p | pregnancy that is observed in fema | ales and can be observed in males | S. |
| Menorrhagia | Mild; iron supplements indicated | Moderate symptoms; medical intervention indicated (e.g., hormones) | Severe; transfusion indicated;<br>surgical intervention indicated<br>(e.g., hysterectomy) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by abnormally heavy vaginal bl | eeding during menses. | | <u> </u> | |
| Nipple deformity | Asymptomatic; asymmetry with slight retraction and/or thickening of the nipple areolar complex | Symptomatic; asymmetry of<br>nipple areolar complex with<br>moderate retraction and/or<br>thickening of the nipple areolar<br>complex | - | - | - |
| Definition: A disorder characteriz | ed by a malformation of the nipple | I | T | Г | |
| Oligospermia | Sperm concentration >48 million/mL or motility >68% | Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Sperm concentration <13<br>million/mL or motility <32% | - | - |
| Definition: A disorder characteriz | red by a decrease in the number of | f spermatozoa in the semen. | 1 | T | |
| Ovarian hemorrhage | Minimal bleeding identified on imaging study or laproscopy; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the ovary. | | | | |
| Ovarian rupture | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by tearing or disruption of the o | varian tissue. | | | |
| Ovulation pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz ovarian follicle. | red by marked discomfort sensation | n in one side of the abdomen betv | veen menstrual cycles, around the | time of the discharge of the ovum | from the |
| Pelvic floor muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles of the pelvic floor. | | | |
| Pelvic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the pelvis. | T | <u> </u> | |
| Penile pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | red by marked discomfort sensation | n in the penis. | ı | <u> </u> | |
| Perineal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the area between the ger | nital organs and the anus. | | |
| Premature menopause | - | - | Present | - | - |
| Definition: A disorder characteriz | ed by ovarian failure before the ag | e of 40. Symptoms include hot fla | shes, night sweats, mood swings | and a decrease in sex drive. | |
| Prostatic hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | Ι - |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by bleeding from the prostate of | gland. | | 1 | 1 |
| Prostatic obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz<br>stream, and incomplete emptying | • • | secondary to enlargement of the p | prostate gland. This results in voidi | ng difficulties (straining to void, sle | ow urine |
| Prostatic pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| D-6-:ki | | instrumental ADL | ADL | | |
| | ed by a sensation of marked disco | | 1 | | 1 |
| Scrotal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the scrotal area. | T | T | 1 |
| Spermatic cord hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the spermation | cord. | • | ' | |
| Spermatic cord obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | 1 | of the contents of the spermatic c | 1 | I | I |
| Testicular disorder | Asymptomatic; clinical or | Symptomatic but not interfering | Severe symptoms; interfering | Life-threatening consequences; | Death |
| TOSTOCIAL GISOTACI | diagnostic observations only; | with urination or sexual | with urination or sexual function; | urgent intervention indicated | Dodin |
| | intervention not indicated | activities; intervention not indicated; limiting instrumental | limiting self care ADL; intervention indicated | | |
| | | ADL | | | |
| Definition: A disorder characteriz | ed by involvement of the testis. | | | I | |
| Testicular hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the testis. | | | | |
| Testicular pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the testis. | 1 | ' | ' |
| Uterine fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | n between the uterus and another | organ or anatomic site. | | • |
| Uterine hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the uterus. | • | • | ' | • |
| Uterine obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | red by blockage of the uterine outle | 1 | 1 . | 1 | 1 |
| Uterine pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | led by a sensation of marked disco | • | ı | 1 | ı |
| Vaginal discharge | Mild vaginal discharge (greater than baseline for patient) | Moderate to heavy vaginal discharge; use of perineal pad | - | - | - |
| | , , | or tampon indicated | | | |
| D C 10 A 10 A 1 A 1 | ed by vaginal secretions. Mucus p | produced by the cervical glands is | discharged from the vagina natura | lly, especially during the childbea | ring years |
| Definition: A disorder characteriz | | | | | |
| Definition: A disorder characteriz | Mild vaginal dryness not interfering with sexual function | Moderate vaginal dryness interfering with sexual function or causing frequent discomfort | Severe vaginal dryness<br>resulting in dyspareunia or<br>severe discomfort | - | - |

| | Rep | productive system and be | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between the vagina and another | organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on<br>clinical exam or imaging study;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema, or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal ulceration; life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation involving the v | agina. Symptoms may include rec | dness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characterize | ed by blockage of vaginal canal. | | 1 | | |
| Vaginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | mfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a rupture in the vaginal wall. | | | | |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or shortening not interfering with physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characterize | ed by a narrowing of the vaginal ca | anal. | | | |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | - | - |
| Definition: A disorder characterize intercourse. | ed by involuntary spasms of the pe | elvic floor muscles, resulting in pa | thologic tightness of the vaginal w | all during penetration such as duri | ng sexual |
| Reproductive system and breast<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adult respiratory distress syndrome | - | - | Present with radiologic findings; intubation not indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterizeurgery. | zed by progressive and life-threater | ning pulmonary distress in the abs | sence of an underlying pulmonary | condition, usually following major t | rauma or |
| Allergic rhinitis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| | zed by an inflammation of the nasa<br>of the sinuses, eyes, middle ear, a | | | - | ay also |
| Apnea | - | - | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | zed by cessation of breathing. | | | I | |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Altered eating habits; coughing or choking episodes after eating or swallowing; medical intervention indicated (e.g., suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or hemodynamic compromise; intubation or urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by inhalation of solids or liquids | s into the lungs. | 1 | | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | zed by the collapse of part or the en | ntire lung. | 1 | T | |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild wheezing); endoscopic evaluation indicated; radiographic evidence of atelectasis/lobar collapse; medical management indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | zed by blockage of a bronchus pas | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | zed by a narrowing of the bronchial | | Covere over-t P. W | Life threater: | Do -# |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | n between a bronchus and the ple | ural cavity. | I | |
| Bronchopulmonary hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g., | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention | Death |

| Respiratory, thoracic and mediastinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| Advance Event | 4 | 2 | | 4 | _ |
| Adverse Event | Mild constant interesting and | 2 | 3 | 4 | 5 |
| Bronchospasm | Mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Limiting self care ADL; oxygen saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a sudden contraction of the | smooth muscles of the bronchial | wall. | | |
| Chylothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thoracentesis or tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charact | erized by milky pleural effusion (abnor | rmal collection of fluid) resulting fr | om accumulation of lymph fluid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription intervention indicated | Moderate symptoms, medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder charact<br>by a distinctive sound. | erized by sudden, often repetitive, spa | asmodic contraction of the thoraci | c cavity, resulting in violent release | e of air from the lungs and usually a | accompar |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an uncomfortable sensation | of difficulty breathing. | | 1 | |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; topical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the nose. | | | | |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe symptoms; interfering with sleep; limiting self care ADL | - | - |
| Definition: A disorder charact | erized by repeated gulp sounds that re | esult from an involuntary opening | and closing of the glottis. This is a | ttributed to a spasm of the diaphra | igm. |
| Hoarseness | Mild or intermittent voice<br>change; fully understandable;<br>self-resolves | Moderate or persistent voice<br>changes; may require<br>occasional repetition but<br>understandable on telephone;<br>medical evaluation indicated | Severe voice changes including predominantly whispered speech | - | - |
| Definition: A disorder charact | erized by harsh and raspy voice arisin | g from or spreading to the larynx. | | | |
| Hypoxia | erized by a decrease in the level of ox | Decreased oxygen saturation with exercise (e.g., pulse oximeter <88%); intermittent supplemental oxygen | Decreased oxygen saturation at<br>rest (e.g., pulse oximeter <88%<br>or PaO2 <=55 mm Hg) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Laryngeal edema | Asymptomatic; clinical or | Symptomatic; medical | Stridor; respiratory distress; | Life-threatening airway | Death |
| | diagnostic observations only; intervention not indicated | intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | hospitalization indicated | compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | erized by swelling due to an excessive | | | | l |
| Laryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube thoracostomy or medical management indicated; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder charact | erized by an abnormal communication | between the larynx and another | organ or anatomic site. | | |
| Laryngeal hemorrhage | Mild cough or trace hemoptysis; laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | erized by bleeding from the larynx. | | | | |
| Definition: A disorder charact | | | 1 | | |

| | Respi | ratory, thoracic and med | iastinai disorders | | |
|---|---|---|---|---|---|
| | | T. | Grade | Г | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngeal mucositis | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered oral intake | Severe pain; severely altered<br>eating/swallowing; medical<br>intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteria | zed by an inflammation involving th | e mucous membrane of the laryn | (. | i - | |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by blockage of the laryngeal ai | rway. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a narrowing of the laryngeal | | | | D " |
| Laryngopharyngeal dysesthesia | n Mild symptoms; no anxiety;<br>intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and swallowing difficulty; limiting self care ADL | Life-threatening consequences | Death |
| Definition: A disorder characteri | zed by an uncomfortable persistent | sensation in the area of the laryn | gopharynx. | | |
| Laryngospasm | - | Transient episode; intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characteri: | zed by paroxysmal spasmodic mus | cular contraction of the vocal cord | ls. | | ' |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hemostasis of bleeding<br>site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri: | ा<br>zed by bleeding from the mediastin | um. | 1/ | l | ı |
| Nasal congestion | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Associated with bloody nasal discharge or epistaxis | - | - |
| | zed by obstruction of the nasal pas | 1 | | | ı |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri. | zed by an abnormal communication | between the pharynx and another | er organ or anatomic site. | I | |
| Pharyngeal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characterize | zed by bleeding from the pharynx. | T | 1 | Γ | |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics indicated; altered oral intake; limiting instrumental ADL | Severe pain; unable to adequately aliment or hydrate orally; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an inflammation involving th | e mucous membrane of the phary | | | ı |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | ized by a necrotic process occurring | in the pharynx. | | | |
| Pharyngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder character | ized by a narrowing of the pharynge | al airway. | , | ' | |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensation | n in the pharyngolaryngeal region. | 1 | i - | , |
| Pleural effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., diuretics or limited therapeutic thoracentesis) | Symptomatic with respiratory<br>distress and hypoxia; surgical<br>intervention including chest tube<br>or pleurodesis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | ized by an increase in amounts of flo | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or associated with pneumothorax; chest tube drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | ized by bleeding from the pleural ca | vity. | | | |
| Pleuritic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensation | n in the pleura. | | <u> </u> | |
| Pneumonitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | ized by inflammation focally or diffus | | | | |
| Pneumothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative intervention indicated; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by abnormal presence of air in | the pleural cavity resulting in the | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | ized by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | |
| Productive cough | 1 | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | - | - |
| | ized by expectorated secretions upo | | Covere diannes er diannes et | Life threatening requireten. | Dooth |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at rest; oxygen indicated; limiting self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder character | ized by accumulation of fluid in the I | ung tissues that causes a disturba | | lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia; radiologic<br>pulmonary fibrosis <25% of lung<br>volume | Moderate hypoxemia; evidence<br>of pulmonary hypertension;<br>radiographic pulmonary fibrosis<br>25 - 50% | Severe hypoxemia; evidence of right-sided heart failure; radiographic pulmonary fibrosis >50 - 75% | Life-threatening consequences<br>(e.g., hemodynamic/pulmonary<br>complications); intubation with<br>ventilatory support indicated;<br>radiographic pulmonary fibrosis<br>>75% with severe<br>honeycombing | Death |
| Definition: A disorder character | ized by the replacement of the lung | tissue by connective tissue, leadir | ng to progressive dyspnea, respira | tory failure or right heart failure. | |
| Pulmonary fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Respi | ratory, thoracic and med | astinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | red by an abnormal communication | between the lung and another or | gan or anatomic site. | I | |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other evaluation | Moderate dyspnea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated<br>with hypoxemia, right heart<br>failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | ed by an increase in pressure with | in the pulmonary circulation due to | lung or heart disorder. | | |
| Respiratory failure | - | - | - | Life-threatening consequences; urgent intervention, intubation, or ventilatory support indicated | Death |
| Definition: A disorder characteriz with an increase in arterial levels | red by impaired gas exchange by t<br>s of carbon dioxide. | he respiratory system resulting in | hypoxemia and a decrease in oxy | genation of the tissues that may be | e associate |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight<br>gain; intervention with fluid<br>restriction and/or diuretics<br>indicated | Moderate signs or symptoms; steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; ventilatory support indicated | Death |
| Definition: A disorder characteriz retinoic acid. | red by weight gain, dyspnea, pleur | al and pericardial effusions, leukoo | cytosis and/or renal failure original | ly described in patients treated wit | h all-trans |
| Sinus disorder | Asymptomatic mucosal crusting; blood-tinged secretions | Symptomatic stenosis or edema/narrowing interfering with airflow; limiting instrumental ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the paranasa | al sinuses. | ' | • | • |
| Sleep apnea | Snoring and nocturnal sleep arousal without apneic periods | Moderate apnea and oxygen<br>desaturation; excessive daytime<br>sleepiness; medical evaluation<br>indicated; limiting instrumental<br>ADL | Oxygen desaturation;<br>associated with hypertension;<br>medical intervention indicated;<br>limiting self care ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by cessation of breathing for sh | nort periods during sleep. | | | |
| Sneezing | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by the involuntary expulsion of | air from the nose. | • | • | |
| Sore throat | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | - | - |
| Definition: A disorder characteriz | ed by of marked discomfort in the | throat | ' | ' | • |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characteriz | red by a high pitched breathing sou | und due to laryngeal or upper airw | ay obstruction. | | |
| Tracheal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characteriz | red by an abnormal communication | between the trachea and anothe | organ or anatomic site. | | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe pain; hemorrhage or respiratory symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an inflammation involving th | | | | I |
| Tracheal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Stridor or respiratory distress<br>limiting self care ADL;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | ed by a narrowing of the trachea. | 1 | • | 1 | ' |

| | Respiratory, thoracic and mediastinal disorders | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Voice alteration | Mild or intermittent change from normal voice | Moderate or persistent change<br>from normal voice; still<br>understandable | Severe voice changes including predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology | - | - |
| Definition: A disorder characteriz | ed by a change in the sound and/o | or speed of the voice. | | | |
| Wheezing | Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe respiratory symptoms<br>limiting self care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a high-pitched, whistling sou | und during breathing. It results from | n the narrowing or obstruction of t | he respiratory airways. | |
| Respiratory, thoracic and mediastinal disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Alopecia | Hair loss of <50% of normal for that individual that is not obvious from a distance but only on close inspection; a different hair style may be required to cover the hair loss but it does not require a wig or hair piece to | piece is necessary if the patient<br>desires to completely<br>camouflage the hair loss; | - | - | - |
| | camouflage | impact | | | |
| Definition: A disorder character | rized by a decrease in density of hair | r compared to normal for a given i | ndividual at a given age and body | location. | |
| Body odor | Mild odor; physician intervention not indicated; self care interventions | Pronounced odor; psychosocial impact; patient seeks medical intervention | - | - | - |
| Definition: A disorder character | rized by an abnormal body smell res | ulting from the growth of bacteria | on the body. | 1 | 1 |
| Bullous dermatitis | Asymptomatic; blisters covering <10% BSA | Blisters covering 10 - 30% BSA;<br>painful blisters; limiting<br>instrumental ADL | Blisters covering >30% BSA;<br>limiting self care ADL | Blisters covering >30% BSA;<br>associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder character | rized by inflammation of the skin cha | racterized by the presence of bull | ae which are filled with fluid. | T | 1 |
| Dry skin | Covering <10% BSA and no associated erythema or pruritus | Covering 10 - 30% BSA and associated with erythema or pruritus; limiting instrumental ADL | Covering >30% BSA and associated with pruritus; limiting self care ADL | - | - |
| Definition: A disorder character | rized by flaky and dull skin; the pores | s are generally fine, the texture is | a papery thin texture. | | |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target lesions covering 10 -<br>30% BSA and associated with<br>skin tenderness | Target lesions covering >30%<br>BSA and associated with oral or<br>genital erosions | Target lesions covering >30%<br>BSA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder character | rized by target lesions (a pink-red rin | g around a pale center). | T | T | |
| Erythroderma | - | Erythema covering >90% BSA without associated symptoms; limiting instrumental ADL | Erythema covering >90% BSA with associated symptoms (e.g., pruritus or tenderness); limiting self care ADL | Erythema covering >90% BSA with associated fluid or electrolyte abnormalities; ICU care or burn unit indicated | Death |
| Definition: A disorder character | rized by generalized inflammatory er | ythema and exfoliation. The inflan | nmatory process involves > 90% o | f the body surface area. | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL | Covering >30% BSA;<br>associated with erythema or<br>tenderness; limiting self-care<br>ADL | - | - |
| Definition: A disorder character | rized by shrinking of adipose tissue. | | 1 | | 1 |
| Hirsutism | In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | - | - | - |
| Definition: A disorder character | rized by the presence of excess hair | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | and under |
| androgen control (beard, mous | • • | | | | |
| Hyperhidrosis | Limited to one site (palms, soles, or axillae); self care interventions | Involving >1 site; patient seeks medical intervention; associated with psychosocial impact | Generalized involving sites<br>other than palms, soles, or<br>axillae; associated with<br>electrolyte/hemodynamic<br>imbalance | - | - |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or<br>density of hair that the patient is<br>either able to camouflage by<br>periodic shaving or removal of<br>hairs or is not concerned | Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) | - | - | - |
| | enough about the overgrowth to use any form of hair removal | plus/minus arms] that requires<br>frequent shaving or use of<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial<br>impact | | | |
| Definition: A disorder characteria | zed by hair density or length beyon | d the accepted limits of normal in | a particular body region, for a part | icular age or race. | |
| Hypohidrosis | - | Symptomatic; limiting instrumental ADL | Increase in body temperature;<br>limiting self care ADL | Heat stroke | Death |
| Definition: A disorder characteri | T . | | | | |
| Lipohypertrophy | Asymptomatic and covering <10% BSA | Covering 10 - 30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% BSA and associated tenderness and narcotics or NSAIDs indicated; lipohypertrophy; limiting self care ADL | - | - |
| Definition: A disorder characteri: | zed by hypertrophy of the subcutan | eous adipose tissue at the site of | multiple subcutaneous injections of | of insulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteria | zed by a change in the color of the | nail plate. | | <b>I</b> | |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the<br>nail bed from the nail plate or<br>nail loss; limiting instrumental<br>ADL | - | - | - |
| Definition: A disorder characteri: | zed by loss of all or a portion of the | nail. | , | • | • |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri: | ा<br>zed by vertical or horizontal ridges | on the nails. | ı | l | Į. |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteria | zed by marked discomfort sensation | n in the skin. | T | Ī | |
| Palmar-plantar<br>erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling,<br>blisters, bleeding, edema, or<br>hyperkeratosis) with pain;<br>limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by redness, marked discomfort | | s of the hands or the soles of the f | eet. | 1 |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | - | - |
| Definition: A disorder characteri. | zed by swelling due to an excessive | e accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Painless erythema and erythema covering <10% BSA | Tender erythema covering 10 - 30% BSA | Erythema covering >30% BSA<br>and erythema with blistering;<br>photosensitivity; oral<br>corticosteroid therapy indicated;<br>pain control indicated (e.g.,<br>narcotics or NSAIDs) | Life-threatening consequences; urgent intervention indicated | Death |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated;<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | - | - |
| Definition: A disorder characterize | zed by an intense itching sensation | | ! | | 1 |
| Purpura Definition: A disorder characteriz | Combined area of lesions covering <10% BSA | Combined area of lesions covering 10 - 30% BSA; bleeding with trauma in and mucous membrane. Newer | Combined area of lesions covering >30% BSA; spontaneous bleeding | -<br>Dider lesions are usually a darker p | -<br>ourple color |
| and eventually become a browni | | | | | |
| Rash acneiform | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder characteriz | zed by an eruption of papules and p | pustules, typically appearing in fac | e, scalp, upper chest and back. | | |
| Rash maculo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering<br>>30% BSA with or without<br>associated symptoms; limiting<br>self care ADL | - | - |
| | zed by the presence of macules (fla<br>upper trunk, spreading centripetally | | nown as morbillform rash, it is one | of the most common cutaneous a | dverse |
| Scalp pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | zed by marked discomfort sensation | n in the skin covering the top and | the back of the head. | ſ | |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA;<br>associated with ulceration | - | - |
| Definition: A disorder characterize | zed by the degeneration and thinning | ng of the epidermis and dermis. | | | |
| Skin hyperpigmentation | Hyperpigmentation covering <10% BSA; no psychosocial impact | Hyperpigmentation covering >10% BSA; associated psychosocial impact | - | - | - |
| Definition: A disorder characterize | zed by darkening of the skin due to | excessive melanin deposition. | | | |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | - | - | - |
| Definition: A disorder characteriz | zed by loss of skin pigment. | | | | |
| Skin induration | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| Definition: A disorder characterize | zed by an area of hardness in the s | kin. | T | Γ | |
| Skin ulceration | Combined area of ulcers <1 cm;<br>nonblanchable erythema of<br>intact skin with associated<br>warmth or edema | Combined area of ulcers 1 - 2<br>cm; partial thickness skin loss<br>involving skin or subcutaneous<br>fat | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to or necrosis of<br>subcutaneous tissue that may<br>extend down to fascia | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or supporting structures with or without full thickness skin loss | Death |
| Definition: A disorder characteriz | zed by circumscribed, inflammatory | and necrotic erosive lesion on the | e skin. | | |
| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | - | - | Skin sloughing covering <10%<br>BSA with associated signs (e.g.,<br>erythema, purpura, epidermal<br>detachment and mucous<br>membrane detachment) | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment) | Death |
| Definition: A disorder characterize | ed by less than 10% total body ski | n area separation of dermis. The | syndrome is thought to be a hyper | sensitivity complex affecting the s | kin and the |
| mucous membranes. | I | | | | 1 |
| Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | - | - | - |
| Definition: A disorder characterize | ed by local dilatation of small vess | els resulting in red discoloration o | f the skin or mucous membranes. | | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characterize | ed by greater than 30% total body | skin area separation of dermis. T | he syndrome is thought to be a hy | persensitivity complex affecting th | e skin and the |
| mucous membranes. | | | | | 1 |
| Urticaria | Urticarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 - 30% BSA; oral intervention indicated | Urticarial lesions covering >30%<br>BSA; IV intervention indicated | - | - |
| Definition: A disorder characterized by an itchy skin eruption characterized by wheals with pale interiors and well-defined red margins. | | | | | |
| Skin and subcutaneous tissue disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Social circumstances | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Menopause | Menopause occurring at age 46 - 53 years of age | Menopause occurring at age 40 - 45 years of age | Menopause occurring before age 40 years of age | - | - |
| Definition: A disorder characteriz | ed by the permanent cessation of | menses, usually defined by 12 co | nsecutive months of amenorrhea i | n a woman over 45 years of age. | |
| Social circumstances - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| procedures - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by leakage of intravascular fluid<br>syndromes, low-flow states, ischel | | | - | |
| failure. | | | | | |
| Flushing | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Symptomatic, associated with hypotension and/or tachycardia; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by episodic reddening of the fa | ce. | | | 1 |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterized by a localized collection of blood, usually clotted, in an organ, space, or tissue, due to a break in the wall of a blood vessel. | | | | | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by an uncomfortable and temp | orary sensation of intense body w | armth, flushing, sometimes accom | panied by sweating upon cooling. | |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic<br>BP 140 - 159 mm Hg or<br>diastolic BP 90 - 99 mm Hg);<br>medical intervention indicated;<br>recurrent or persistent (>=24<br>hrs); symptomatic increase by<br>>20 mm Hg (diastolic) or to | Stage 2 hypertension (systolic<br>BP >=160 mm Hg or diastolic<br>BP >=100 mm Hg); medical<br>intervention indicated; more<br>than one drug or more intensive<br>therapy than previously used<br>indicated | Life-threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit, hypertensive<br>crisis); urgent intervention<br>indicated<br>Pediatric: Same as adult | Death |
| Definition: A disorder characterist | zed by a pathological increase in bl | >140/90 mm Hg if previously WNL; monotherapy indicated Pediatric: recurrent or persistent (>=24 hrs) BP >ULN; monotherapy indicated | Pediatric: Same as adult | og 140 over 90 mm Hg | |
| Hypotension | Asymptomatic, intervention not | Non-urgent medical intervention | · | Life-threatening and urgent | Death |
| riypotonolori | indicated | indicated | hospitalization indicated | intervention indicated | Bouii |
| Definition: A disorder characterization | zed by a blood pressure that is belo | ow the normal expected for an indi | ividual in a given environment. | | |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by the loss of lymph fluid into the | 1 | Ĺ | 1 | 1 |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery<br>skin texture; papillary formation;<br>limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by excessive fluid collection in | tissues that causes swelling. | | T | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characteriz | zed by a cystic lesion containing ly | mph. | | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of<br>ischemia managed non-<br>surgically and without<br>permanent deficit | Recurring or prolonged (>=24<br>hrs) and/or invasive intervention<br>indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characterize | zed by impaired circulation to an ex | ctremity. | 1 | 1 | |
| Phlebitis | - | Present | - | - | - |
| | zed by inflammation of the wall of a | vein. | | | |
| Superficial thrombophlebitis Definition: A disorder characterize | -<br>zed by a blood clot and inflammatio | 1 | l -<br>e extremities. | 1- | 1 - |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences; urgent multi-modality intervention indicated (e.g., lysis, thrombectomy, surgery) | Death |
| Definition: A disorder characterized by obstruction of the blood flow in the superior vena cava. Signs and symptoms include swelling and cyanosis of the face, neck, and upper arms, | | | | | |
| cough, orthopnea and headache | | | | | |
| Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | Thrombosis (e.g., uncomplicated pulmonary embolism [venous], non-embolic cardiac mural [arterial] thrombus), medical intervention indicated | Life-threatening (e.g., pulmonary embolism, cerebrovascular event, arterial insufficiency); hemodynamic or neurologic instability; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream. | | |
| Vasculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the w | rall of a vessel. | • | • | |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of ischemia managed medically and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a decrease in blood supply | due to narrowing or blockage of a | visceral (mesenteric) artery. | | |
| Vascular disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |







NIH Publication No. 09-5410 Revised June 2010 Reprinted June 2010



# Appendix B: Pemphigus Disease Area Index (PDAI)

### Pemphigus Disease Area Index (PDAI)

| Skin | Activity | | Damage Post-inflammatory |
|---|---|---|---|
| Anatomical Locatio | Erosion/Blisters or new erythem | sion/Blisters or new erythema | |
| | absent 1-3 lesions, up to one >2 cm in any diameter, none > 6 cm 2-3 lesions, at least two > 2 cm diameter, none > 6 cm 3 >3 lesions, none > 6 cm diameter 5 >3 lesions, and/or at least one >6 cm 3 lesions and/or at least one lesion >16 cm diameter or entire area | Number<br>lesions if<br>≤ 3 | from resolving lesion 0 absent 1 present |
| Ears | | | |
| Nose | | | |
| Rest of the face | | | |
| Neck | | | |
| Chest | | | |
| Abdomen | | | |
| Back, buttocks | | | |
| Arms | | | |
| Hands | | | |
| Legs | | | |
| Feet | | | H |
| Genitals | | | 40 |
| Total skin | /120 | | /12 |
| Scalp | | | |
| Scalp | Erosion/Blisters or new erythem | а | Post-inflammatory<br>hyperpigmentation or erythen<br>from resolving lesion |
| | 0 absent 1 in one quadrant 2 two quadrants 3 three quadrants 4 affects whole skull 10 at least one lesion > 6 cm | | 0 absent<br>1 present |
| Total Scalp (0-10) | /10 | | /1 |
| Mucous mer | nbrane | | |
| Anatomical<br>Location | Erosion/Blisters | | |
| | 0 absent<br>1 1 lesion<br>2 2-3 lesions<br>5 >3 lesions or 2 lesions >2 cm<br>10 entire area | Number<br>lesions<br>if ≤ 3 | |
| Eyes | | | |
| Nose | | | |
| Buccal mucosa | | | |
| Hard palate | | | |
| Soft palate | | | |
| Upper gingiva | | | |
| Lower gingiva | | | |
| Tongue | | $\vdash$ | |
| | I | ı I | |
| Floor of mouth | | - | |
| Labial bucosa | | | |
| Labial bucosa<br>Posterior pharynx | | | |
| Labial bucosa | /120 | | |

Copyright ©2007 University of Pennsylvania; All Rights Reserved.

# Syntimmune, Inc.

### SUMMARY OF CHANGES TO CLINICAL STUDY PROTOCOL

# A Phase 1b, Multicenter, Open-Label, Safety, Tolerability, and Activity Study of SYNT001 in Subjects with Chronic Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**IND Number:** 132727

Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

257 Park Avenue South

15th Floor

New York, NY 10010

Medical Monitor:

Wallace House

17-21 Maxwell Place Stirling, Scotland FK81JU

Mobile Phone: PPD

Office Phone: PPD

ext. PPD

Original Protocol:19 December 2016Amendment 1.118 January 2017Amendment 2.012 April 2017Amendment 3.010 October 2017

### **Confidentiality Statement**

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. and any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

#### **SUMMARY**

The SYNT001-103 protocol has been amended under version 3.0 as follows:

- Medical Monitor and emergency contact information has been updated
- Clarification of allowable corticosteroids
- Additional exploratory biomarker and subsequent increase in total blood volume included
- Increase maximum BMI from 35.0 to 39.9 mg/m<sup>2</sup>
- Allowance of urine or serum pregnancy tests for women of childbearing potential at screening
- Clarification of the restriction on cellular therapy
- Provide guidance on the use of premedications for SYNT001 dosing
- Clarification of the type of skin the optional biopsies may be taken from
- Clarification of the method of sample collection for FCGR2A
- Clarification of the treatment for the single Grade 2 AE in the Phase 1a study
- Clarification of the data collected as part of the patient relevant medical history
- Removal of RR Interval as a required part of the ECG assessments
- Clarification that subjects exceeding a specific weight are not to be enrolled into the 30 mg/kg or higher dose groups based on theoretical host cell DNA levels per dose
- Clarification for the management of a Grade 1 infusion reaction.
- Provides a maximum duration of infusion in accordance with the requirements for SYNT001 preparation and administration outlined in the pharmacy manual
- Clarification of SAE reporting requirements and IRB notifications
- Sponsor contact information has been updated
- Various typographical and formatting corrections as well as corrections for consistency made throughout the document.

Syntimmune, Inc.  10 October 2017

### **SPECIFIC CHANGES**

Text deletions are shown using strike through font; new text added in *italic font*. Listed page numbers are based on Protocol Amendment 2.0, dated 12 April 2017.

| | ction, Page<br>Number | | Original Text | Revised Text | Rationale |
|---|---|---|---|---|---|
| Cover, | page 1 | Blythe Tl | nomson, MD | Richard Kay, MD | Medical Monitor information updated |
| | | | PP PP reet, | Wallace House | |
| | D D | Cambridg | D D 01240 | 17-21 Maxwell Place | |
| | | | | Stirling, Scotland FK81JU | |
| | | | | Mobile Phone: (+44) 7747 621 827 | |
| | | PP<br>D | | Office Phone: (+44) 1786 460 400 ext. | |
| PP | | PP | | 24461 | |
| EmeD | cy Contact | BlyD | om , MD | Richard Kay, MD | Medical Monitor information updated |
| Info | tion, page 3 | b.tl | @medpace.com | _r.kay@medpace.com | |
| | | Μc | one: 1-513-748-2122 | Mobile phone: (+44) 7747 621 827 | |
| | | PP<br>D | ne: 1-PP -579-9911 ext. | Office phone: (+44) 1786 460 400 ext. | |
| | | | | 24461 | |
| Synops | | | | Exploratory biomarkers to | Added an additional exploratory objective to |
| Explor | • | | | investigate immune response | investigate other possible biomarkers associated |
| Objecti | ives, page 7 | | | associated with pemphigus | with the pemphigus immune response |
| Synops | sis, Diagnosis | c. If bein | PP PP d with corticosteroids, | c. If being treated with corticosteroids, | Clarification of allowable corticosteroids |
| and ma | in entry | dose mp | D mg/kg/day and stable | dose must be $\leq 1 \text{mg/kg/day } of$ | |
| | , page 9 | (< 10 n) | n dose) for 2 weeks | prednisone or equivalent and stable (< | |
| PP<br>D | | pri | g | 10% change in dose) for 2 weeks prior | |
| | | | | to screening | |
| Sync | s, Diagnosis | 5. | ass index (BMI) 18.5 – 35.0 | 5. Body mass index (BMI) 18.5 – | Patients who may be otherwise eligible to |
| and | entry | kg/ | | 39.9 <del>35.0 kg</del> /m <sup>2</sup> ; | participate in the study are excluded due to BMI. |
| crite | page 9 | | PP | | We would like to be able to offer these |
| | | | D | | individuals the opportunity to participate |
| - | s, Diagnosis | 6. | egativ rine pregnancy test | 6 Has a negative <del>urine pregnancy test</del> | Allows for serum or urine tests as per |
| | in entry | * | en of childbearing potential) | (for women of childbearing potential) | institutional standards |
| criteria | , page 9 | | ted prior to the first dose of | documented prior to the first dose of | |
| | | study dru | <u> </u> | study drug; | |
| | is, Diagnosis | 10. Cellu | lar therapy at any time prior | 10. Cellular therapy, <i>including CAR-T</i> , | To further clarify the restriction on all cellular |
| | in entry | to screen | ing | therapy at any time prior to screening | therapy |
| criteria | , page 10 | | | | |

Syntimmune, Inc.  10 October 2017


| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Synopsis, Prohibited Concomitant Treatments, page 11 | All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. | All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. Premedication is discouraged as prophylaxis against AEs or infusion reactions unless medically indicated from either past medical history, prior infusion reactions or AEs resulting from SYNT001 infusions. | Infusion reactions are a common adverse effect of IV administration of some, but not all monoclonal antibodies (mAb). Infusion reactions most commonly occur with the first infusion and are often related to the infusion rate. For mAbs with frequent infusion reactions, it is recommended that pre-medications, such as corticosteroids, acetaminophen and/or antihistamines, are administered prior to infusion, especially with the first infusion. However, pre-medications are generally not recommended for mAbs associated with no or mild infusion reactions. No infusion reactions occurred in the recently completed healthy volunteer phase 1a single-ascending dose study, where infusions were given over 1 hour at doses up to 30 mg/kg. As such, Syntimmune does not currently believe that it is necessary or appropriate to administer pre-medications to patients who will be receiving SYNT001 at the same doses and infusion rate as in the phase 1a study. If frequent infusion reactions are observed in the phase 1b study, the issue of pre-medication will be revisited. |

| Section, Page | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Number | | | |
| Pharmacodynamics/ | PD samples will be collected for | PD samples will be collected for | Added an additional exploratory objective to |
| Activity, page 13 | analysis of IgG (serial assessment of | analysis of IgG (serial assessment of | investigate other possible biomarkers associated |
| | IgG levels to identify Cmin, Tmin); | IgG levels to identify Cmin, Tmin); | with the pemphigus immune response |
| | IgG1-4 subtype levels; IgA levels; IgM | IgG1-4 subtype levels; IgA levels; IgM | |
| | levels; albumin levels; anti-Dsg (1 and | levels; albumin levels; anti-Dsg (1 and | |
| | 3) antibody levels; serum AECA by | 3) antibody levels; serum AECA by | |
| | direct immunofluorescence; CIC; C3; | direct immunofluorescence; CIC; C3; | |
| | exploratory biomarkers (FCGR2A | exploratory biomarkers (FCGR2A | |
| | SNP, RNAseq, urine IgG, CD3+CD4+ | SNP, RNAseq, urine IgG, CD3+CD4+ | |
| | T, CD3+CD8+ T, monocytes, NK cells | T, CD3+CD8+ T, monocytes, NK cells | |
| | and B cells). | and B cells) and additional exploratory | |
| | | analyses to investigate immune | |
| | | response associated with pemphigus. | |
| Synopsis, Skin | Optional skin biopsy samples will be | Optional skin biopsy samples from | Clarifies type of skin the optional biopsies may |
| Biopsy, page 13 | collected on Day 0 pre-dose and on | lesional or non-lesional skin will be | be taken from |
| | Days 1, 2, 14, 33, 56 and 84 to analyze | collected on Day 0 pre-dose and on | |
| | SYNT001 levels. | Days 1, 2, 14, 33, 56 and 84 to analyze | |
| | | SYNT001 levels. | |
| Criteria for | | • Exploratory biomarkers to investigate | Added an additional exploratory objective to |
| Evaluation, page 14 | | immune response associated with | investigate other possible biomarkers associated |
| | | pemphigus | with the pemphigus immune response |
| Table 1, Study | | Pemphigus immune response | Sample collection for exploratory pemphigus |
| Assessments, page 16 | | biomarkers | immune response biomarkers added at Days 0, |
| | | | 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84 and 112 |
| Table 1, Study | FCGR2A <sup>m</sup> | FCGR2A <sup>m</sup> by buccal swab | Clarifies method of sample collection |
| Assessments, page 16 | | | |
| Table 1, Study | m: Samples to be collected and stored; | m: Buccal Samples to be collected | Clarifies method of sample collection |
| Assessments, page 17 | pending review of clinical and | and stored; pending review of clinical | |
| | pharmacodynamics assessments | and pharmacodynamics assessments | |

| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Section 2.2, Selection | No AEs were observed in the 1 and 3 | No AEs were observed in the 1 and 3 | Clarifies that no treatment was given for the |
| of Doses in this | mg/kg dose cohorts. A single Grade 2 | mg/kg dose cohorts. A single Grade 2 | Grade 2 AE of headache in the Phase 1a study. |
| Study, page 27 | AE was observed; a headache in the 10 | AE was observed; a headache in the 10 | - |
| | mg/kg cohort., treated with | mg/kg cohort-treated with | |
| | acetaminophen. | acetaminophen | |
| Section 3.3, | | o Exploratory biomarkers to | Added an additional exploratory objective to |
| Exploratory | | investigate immune response associated | investigate other possible biomarkers associated |
| Objectives, Page 29 | | with pemphigus | with the pemphigus immune response |
| Section 4.2, | | • Exploratory biomarkers to investigate | Added an additional exploratory objective to |
| Exploratory Outcome | | immune response associated with | investigate other possible biomarkers associated |
| Measures, page 31 | | pemphigus | with the pemphigus immune response |
| Section 5.2, Inclusion | c. If being treated with corticosteroids, | c. If being treated with corticosteroids, | Clarification of allowable corticosteroids |
| Criteria, page 34 | dose must be $\leq 1 \text{mg/kg/day}$ and stable | dose must be $\leq 1 \text{mg/kg/day } of$ | |
| | (< 10% change in dose) for 2 weeks | prednisone or equivalent and stable (< | |
| | prior to screening | 10% change in dose) for 2 weeks prior | |
| | | to screening | |
| Section 5.2, Inclusion | 5. Body mass index (BMI) 18.5 – 35.0 | 5. Body mass index (BMI) 18.5 – | Patients who may be otherwise eligible to |
| Criteria, page 35 | kg/m2; | <i>39.9</i> <del>35.0</del> kg/m2; | participate in the study are excluded due to BMI. |
| | | | We would like to be able to offer these |
| | | | individuals the opportunity to participate |
| Section 5.2, Inclusion | 6. Has a negative urine pregnancy test | 6. Has a negative urine pregnancy test | Allows for serum or urine tests as per |
| Criteria, page 35 | (for women of childbearing potential) | (for women of childbearing potential) | institutional standards |
| | documented prior to the first dose of | documented prior to the first dose of | |
| | study drug; | study drug; | |
| Section 5.3, | 10. Cellular therapy at any time prior | 10. Cellular therapy, including CAR-T, | To further clarify the restriction on all cellular |
| Exclusion Criteria, | to screening | at any time prior to screening | therapy |
| page 36 | | | |

| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Section 6.2, Demographics and Medical History, page 37 | Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and eCRF. Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery, transfusions and concomitant treatments. | Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and eCRF. Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery, transfusions and concomitant treatments, including relevant clinical response to past disease specific treatments and duration as well as dosing of such treatments. | Clarifies data collected as part of the patient relevant medical history |
| Section 6.6, 12-Lead<br>Electrocardiogram<br>(ECG), page 38 | The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant. | The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant. | Not all study sites have ECG machines that report the RR interval. As heart rate is already being collected as part of clinical evaluation of vital signs, this measure does not provide additional information. ECG machines do provide an estimated heart rate over a 10-second recording and this is a more clinically meaningful outcome measure. |
| Section 6.7, Clinical<br>Laboratory<br>Measurements, page<br>39 | The total blood draw for each subject who completes the study at Day 112, will be approximately 381 mL. | The total blood draw for each subject who completes the study at Day 112, will be approximately 381-433 mL. | Increase due to additional sample collection |
| Section 6.7.5, Table<br>4, Pharmacodynamic<br>Sampling, page 42 | Exploratory biomarker (FCGR2A SNP) | • Exploratory biomarker (FCGR2A SNP, via buccal swab) | Clarifies method of sample collection |

| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Section 6.7.5, Table<br>4, Pharmacodynamic<br>Sampling, page 42 | | • Exploratory pemphigus immune response Days, 0, 7, 14, 21, 28, 33, 42, 56, 84, 112 | Sample collection for exploratory pemphigus immune response biomarkers added at Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84 and 112 |
| Section 6.9, Prior and<br>Concomitant<br>Medications, page 43 | All medications a subject receives within 14 days prior to enrollment through the end of the study will be documented on the source document and eCRF. | All medications a subject receives within 14 days prior to enrollment through the end of the study will be documented on the source document and eCRF. A history of treatments taken for primary disease, even if not taken within the 14 days prior to enrollment, will be collected. | Clarifies data collected as part of the patient relevant medical history |
| Section 6.12, Skin<br>Biopsy, page 44 | Optional skin biopsy samples will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33, 56 and 84 to analyze SYNT001 levels | Optional skin biopsy samples <i>from lesional or non-lesional skin</i> will be collected on Day 0 pre-dose and on Days 1, 2, 14, 33, 56 and 84 to analyze SYNT001 levels | Clarifies type of skin biopsies may be taken from |
| Section 7.2,<br>Enrollment and First<br>Treatment: Dose 0,<br>page 46 | • FCGR2A SNP | FCGR2A SNP via buccal swab | Clarifies method of sample collection |
| Section 7.2,<br>Enrollment and First<br>Treatment: Dose 0,<br>page 46 | | Exploratory pemphigus immune<br>response biomarkers | Added an additional exploratory objective to investigate other possible biomarkers associated with the pemphigus immune response |
| Section 7.5, Follow-<br>up Day 5, page 48 | | Exploratory pemphigus immune<br>response biomarkers | Added an additional exploratory objective to investigate other possible biomarkers associated with the pemphigus immune response |
| Section 7.6,<br>Treatment Day 7<br>(Dose 2), page 48 | | Exploratory pemphigus immune<br>response biomarkers | Added an additional exploratory objective to investigate other possible biomarkers associated with the pemphigus immune response |

Syntimmune, Inc.  10 October 2017

| Section, Page<br>Number | Original Text | | Revised Text | Rationale |
|---|---|---|---|---|
| Section 7.7, Dose 2 | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| Follow-up Day 12, | | | response biomarkers | investigate other possible biomarkers associated |
| page 49 | | | | with the pemphigus immune response |
| Section 7.8, | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| Treatment Day 14 | | | response biomarkers | investigate other possible biomarkers associated |
| (Dose 3), page 50 | | | | with the pemphigus immune response |
| Section 7.9, Dose 3 | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| Follow-up Day 19, | | | response biomarkers | investigate other possible biomarkers associated |
| page 51 | | | | with the pemphigus immune response |
| Section 7.10, | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| Treatment Day 21 | | | response biomarkers | investigate other possible biomarkers associated |
| (Dose 4), page 51 | | | | with the pemphigus immune response |
| Section 7.11, | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| Treatment Day 28 | | | response biomarkers | investigate other possible biomarkers associated |
| (Dose 5), page 52 | | | | with the pemphigus immune response |
| Section 7.14, Follow- | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| up Day 33, page 54 | | | response biomarkers | investigate other possible biomarkers associated |
| | | | | with the pemphigus immune response |
| Section 7.15, Follow- | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| up Day 42, page 55 | | | response biomarkers | investigate other possible biomarkers associated |
| | | | | with the pemphigus immune response |
| Section 7.16, Follow- | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| up Day 56, page 56 | | | response biomarkers | investigate other possible biomarkers associated |
| | | | | with the pemphigus immune response |
| Section 7.17, Follow- | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| up Day 84, page 56 | | | response biomarkers | investigate other possible biomarkers associated |
| | | | | with the pemphigus immune response |
| Section 7.18, Follow- | | • | Exploratory pemphigus immune | Added an additional exploratory objective to |
| up Day 112, page 57 | | | response biomarkers | investigate other possible biomarkers associated |
| | | | | with the pemphigus immune response |

| Section, Page | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Number | | | |
| Section 9.1,<br>SYNT001, page 61 | The specification for host cell DNA in SYNT001 is < 2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing is limited to 5000 mg SYNT001. Therefore, at the highest dose possible in this study (45 mg/kg), maximum subject weight will be limited to 111 kg. | The specification for host cell DNA in SYNT001 is < 2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing is limited to 5000 mg SYNT001. Therefore, the maximum subject weight allowed for enrollment into the 30 mg/kg dose cohort is 166 kg and the maximum subject weight allowed for enrollment into the highest dose possible in this study (45 mg/kg), maximum subject | Clarifies that subjects exceeding a specific weight are not to be enrolled into the 30 mg/kg or higher dose groups based on theoretical host cell DNA levels per dose. |
| | | weight will be limited to is 111 kg. | |

| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Section 9.6.1,<br>Infusion Reaction,<br>page 63 | Management of Grade 1 infusion reactions include decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen. Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. See Figure 1 and Figure 2 for details on the management of Grades 1- 2 and Grade 3 infusion reactions. The severity of and management of allergic or infusion-related reactions will be graded and managed using NCI CTCAE Version 4.03 (see Table 5). | Management of Grade 1 infusion reactions include <i>interrupting the infusion or</i> decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone or acetaminophen, <i>either alone or in combination, depending on the subject's signs and symptoms. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 administration. Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. See Figure 1 and Figure 2 for details on the management of Grades 1– 2 and Grade 3 infusion reactions. The severity of and management of allergic or infusion-related reactions will be graded and managed using NCI CTCAE Version 4.03 (see Table 5).</i> | Provides clarification for the management of a Grade 1 infusion reaction. Provides a maximum duration of infusion in accordance with the requirements for SYNT001 preparation and administration outlined in the pharmacy manual. |
| Section 9.6.1, Figure 1 Title, page 64 | Management of Mild (Grade 1) to<br>Moderate (Grade 2) Infusion Reactions | Management of Mild (Grade 1) to Moderate (Grade 2) Infusion Reaction | To be consistent with prior section regarding management of a Grade 1 infusion reaction and with CTCAE v4.03 definition of a Grade 1 infusion reaction. |

| Section, Page | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Number | | | |
| Section 9.6.1, Figure | Consider pre-medicating the subject | Consider pre-medicating the subject | Provision of a maximum duration of infusion in |
| 1, last box, page 64 | with the same medication(s) 20-30 | with the same medication(s) 20-30 | accordance with the requirements for SYNT001 |
| | minutes in advance of subsequent | minutes in advance of subsequent | preparation and administration as outlined in the |
| | administrations of SYNT001 and | administrations of SYNT001 and | pharmacy manual. |
| | starting infusion at 50% of the planned | starting infusion at 50% of the planned | |
| | infusion rate for the first 30 minutes, | infusion rate for the first 30 minutes, | |
| | then returning to the intended infusion | then returning to the intended infusion | |
| | rate in the absence of any infusion | rate in the absence of any infusion | |
| | reaction | reaction. If the infusion is interrupted | |
| | | or the infusion rate is decreased, it is | |
| | | important to note that all study drug | |
| | | infusions must be completed within 4 | |
| | | hours of SYNT001 administration. | |

| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Section 10, Concomitant Medication and Treatment, page 69 | All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. | All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not excluded below. Topical antibiotics are permitted to treat active infections that occur on study. Topical or systemic treatments for oral candidiasis are permitted. Topical lidocaine for transient pain relief is acceptable as needed. Significant increases in anti-pemphigus medications will result in subjects being discontinued from the study. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study are permitted. Premedication is discouraged as prophylaxis against AEs or infusion reactions unless medically indicated from either past medical history, prior infusion reactions or AEs resulting from SYNT001 infusions. | Infusion reactions are a common adverse effect of IV administration of some, but not all monoclonal antibodies (mAb). Infusion reactions most commonly occur with the first infusion and are often related to the infusion rate. For mAbs with frequent infusion reactions, it is recommended that pre-medications, such as corticosteroids, acetaminophen and/or antihistamines, are administered prior to infusion, especially with the first infusion. However, pre-medications are generally not recommended for mAbs associated with no or mild infusion reactions. No infusion reactions occurred in the recently completed healthy volunteer phase 1a single-ascending dose study, where infusions were given over 1 hour at doses up to 30 mg/kg. As such, Syntimmune does not currently believe that it is necessary or appropriate to administer pre-medications to patients who will be receiving SYNT001 at the same doses and infusion rate as in the phase 1a study. If frequent infusion reactions are observed in the phase 1b study, the issue of pre-medication will be revisited. |

| Section, Page<br>Number | Original Text | Revised Text | Rationale |
|---|---|---|---|
| Section 11.3.9.1,<br>Governing<br>Regulatory<br>Requirements, page<br>76 | Written submission must be made by the sponsor to the FDA and the IRBs as soon as possible and in no event later than 15 calendar days after the sponsor's initial notification of the event. The sponsor shall also inform all Investigators. | Written submission must be made by the sponscPP the F PPD the IRBs as vePP ater that ca PP spo 's D n o eve Th PPD sti | Clarifies that notification to IRBs is not a responsibility of the sponsor. |
| Section 11.3.9.2,<br>Time Frame for<br>Reporting, page 76 | Any death, SAE, pregnancy, or unexpected (and severe) AE experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the sponsor (or designee). | rmed consent the last study trong, must be promptly reported (within 24 hours of the Investigator becoming awpper telephons of the Investigator becoming awpper the proper the proper the proper to the proper the proper to the p | Clarifies that adverse (severe) events that are not considered SAEs do not need to be reported within 24 hours but reported per section 11.3.6. |
| Section 11.3.9.2,<br>Time Frame for<br>Reporting, page 77 | Medical Safety Contact | Me 1S | Medical Monitor information updated |
| Section 14, Study<br>Administration,<br>Table 6, page 86 | Sponsor Contact: Ryan Iarrobino SVP Clinical Operations and Data Management Phone: 617-913-1681 Email: ryan@syntimmune.com | nsor Contact: Ry SVP Clinical Operations and Data Management Phone: 617-913-1681 Email: ryan@syntimmune.com | Sponsor contact information updated |

| Section, P<br>Numbe | _ | | Original Text | | Revised Text | Rationale |
|---|---|---|---|---|---|---|
| Section 14,PP | dy | | Sponsor Medical Direc | ctor: | Sponsor Contact and Medical Director: | Sponsor contact information updated |
| AdministraD | , | | Laurence Blumberg, M | <b>I</b> D | Laurence Blumberg, MD | |
| Table 6, pa | 6 PP | | Founder and Chief Op | erating Officer | President and Chief Operating Officer | |
| | D | | Phone: 917-4-22PP | | Phone: 917-415-2210 | |
| PP | | | Email: laur D nti D | ne.com | Email: laur@syntimmune.com | |
| Section | PP | | Blythe Thom | | Richard Kay, MD | Medical Monitor information updated |
| Admini | D | PP | Medpace | | Medpace | |
| Table 6 | | D | 43 Thorndike ee | | Wallace House | |
| | | | Cambridge, 01 | | 17-21 Maxwell Place | |
| | | | | xt.27201 | Stirling, Scotland FK81JU | |
| | | | Email: b.thoms PP m | edpace.com | Phone: (+44) 1786 460 400 extension | |
| | | | J | | 24461 | |
| | | | Email: r.kay@medpace.com | | | |



# SYNTIMMUNE

02-Mar-2018

**Protocol Number:** 

SYNT001-103

**IND Number:** 

132727

**Study Drug:** 

SYNT001

**Protocol Version, Date:** 

3.0 dated 10-October-2017

Clarification Letter Version: 4.0

Subject:

**Sponsor Medical Director** 

The purpose of this memo is to update the Medical Director details and contact information. Deleted text is crossed through and new text is in italics.

This text will be formally revised in the next forthcoming protocol amendment.

### **Section 14.1 (page 86)**

### **Current Text:**

**Table 1:** Study Administrative Structure



271 Waverley Oaks Road, Suite 104, Waltham, MA 02452

Page 1 of 2

Sincerely,

Sphanie Valler

Stephanie Haller

Vice President, Clinical Operations

Syntimmune, Inc.

DDD

# SYNTIMMUNE, INC. CLINICAL STUDY PROTOCOL

A Phase 1b/2, Multicenter, Open-Label, Safety, and Dose-Finding Study of SYNT001 in Subjects with Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

IND Number: 132727 Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

116 Huntington Avenue

Suite 301

Boston, MA 02116

Medical Monitor:

Wallace House

17-21 Maxwell Place Stirling, Scotland FK81JU

Mobile Phone: PPD Office Phone: PPD

ext. PPD

Original Protocol:18 January 2017Amendment 1.1:21 March 2017Amendment 2.012 April 2017Amendment 3.010 October 2017Amendment 4.08 June 2018

### CONFIDENTIALITY STATEMENT

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. Any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

### SPONSOR SIGNATURE

I have read and approve this protocol. My signature, in conjunction with the signature of the Investigator, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP), the United States Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| PPD | 8 JUNE 2018 |
|------------------|-------------------|
| | Date of Signature |
| Syntimmune, Inc. | |

### **INVESTIGATOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the Sponsor, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP), the United States Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| Nothing in this document is intended to limit the authority of a physician to provide emergency medical care under applicable regulations. | |
|---|---|
| Investigator Signature | Date of Signature |
| Name of Investigator (please print) | |

## 1. SYNOPSIS

| Study title | A Phase 1b/2, Multicenter, Open-Label, Safety, and Dose-Finding Study of SYNT001 in Subjects with Pemphigus (Vulgaris or Foliaceus) |
|---|---|
| Sponsor | Syntimmune, Inc. |
| Protocol number | SYNT001-103 |
| Clinical phase | Phase 1b/2 |
| Number of study centers | Approximately 10 global study sites |
| Study rationale | Pemphigus is a potentially life-threatening group of rare blistering autoimmune diseases that affect the skin and mucous membranes. The exact cause is unknown, though autoantibodies are thought to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. The prognosis of pemphigus has markedly improved over the last decades with the prognosis of pemphigus are profiled to a profiled the prognosis of pemphigus has markedly improved over the last decades with |
| | steroid therapy. Nevertheless, mortality remains an issue (1.6% to 12% of cases) (Hsu et al., 2016; Kasperkiewicz et al., 2017; Langan et al., 2008). In these cases, death typically occurs as a consequence of treatment-related systemic infections and in a smaller proportion, as a consequence of superinfected lesions. While steroids have greatly improved patient outcomes, they are associated with serious and long-lasting side effects; therefore, their use should be limited as much as possible. Although other currently available treatments for certain autoimmune disorders, including immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they can be associated with significant adverse effects and delayed or non-durable responses. |
| | SYNT001 targets key mechanisms contributing to pathology in a variety of immunoglobulin G (IgG)-mediated autoimmune disorders. When administered to healthy subjects, SYNT001 has been shown to significantly decrease total IgG, as well as immune complexes with which IgG is associated. Based on these results, it is predicted that SYNT001 will also reduce the levels of pathogenic autoantibodies. This could lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for sustained disease modification. Thus, this study is being conducted to evaluate the safety and immunogenicity and determine a minimally effective dose (MED) of intravenous (IV) SYNT001 in pemphigus patients. |
| Study objectives and endpoints | The study objectives and their corresponding endpoints (primary, secondary, and exploratory) are detailed below. |

| <b>Primary Objectives</b> | Primary Endpoints |
|---|---|
| Safety: To evaluate the safety of once-weekly IV infusions of SYNT001 at different dose levels and dosing durations in subjects with pemphigus (vulgaris or foliaceus) | Safety: The evaluation of SYNT001 safety based on vital signs, physical examinations, electrocardiograms (ECGs), clinical safety laboratory tests, the incidence of adverse events (AEs), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) summarized by cohort, severity, and relationship to study product |
| Dose Selection: To determine a MED of SYNT001 as assessed by (i) total IgG level nadir and (ii) the proportion of subjects that meet the criteria for response by Pemphigus Disease Area Index total activity score (PDAI) | Dose Selection: The determination of dose and dosing duration of SYNT001 that achieves (i) total IgG level nadir decrease by ≥60% and ≤90% from baseline and (ii) a PDAI total activity score of ≥50% reduction from baseline to allow further clinical development in subjects with pemphigus (vulgaris or foliaceus) |
| Secondary Objectives | Secondary Endpoints |
| To determine the pharmacokinetics (PK) of SYNT001 following onceweekly IV infusions at different dose levels and dosing durations | The determination of PK parameters including half-life $(t_{1/2})$ , maximum serum concentration determined directly from the concentration-time profile $(C_{max})$ , observed time of peak plasma concentration $(T_{max})$ , area under the serum concentration-time curve from pre-dose $(time_0)$ to 24 hours post-dose $(AUC_{0-24})$ , and area under the serum concentration-time curve from pre-dose $(time_0)$ to infinity $(AUC_{0-\infty})$ , $(Cohort\ 1)$ ; maximum plasma concentration determined directly from the concentration-time profile $(C_{max})$ and $T_{max}$ $(Cohort\ 2$ onwards) summarized by cohort and timepoint |
| To evaluate the effect of once-<br>weekly doses of SYNT001 at<br>different dose levels and dosing<br>durations on pharmacodynamics<br>(PD) biomarkers | The evaluation of PD biomarkers based on absolute serum levels and percent change from baseline in serum levels of total immunoglobulin G (IgG), IgG subtypes (IgG1-4), immunoglobulin A (IgA), immunoglobulin M (IgM), albumin, and CIC summarized by cohort and timepoint |

| T= | |
|---|---|
| To assess the effect of once-weekly doses of SYNT001 at different dose levels and dosing durations on disease markers | <ul> <li>The assessment of pemphigus disease activity by responses on PDAI based on absolute and percent change from baseline will be summarized by cohort and timepoint.</li> <li>The assessment of pemphigus disease pathogenic antibody levels based on absolute and percent change from baseline of serum anti-desmoglein 1 and 3 antibody (anti-Dsg 1 and anti-Dsg 3) levels that will be summarized by cohort and timepoint</li> </ul> |
| To measure the immunogenicity of once-weekly administered SYNT001 at different dose levels and dosing durations | The immunogenicity of once-weekly administered SYNT001 as determined by presence of anti-SYNT001 binding antibodies and neutralizing antibodies summarized by cohort and timepoint |
| <b>Exploratory Objectives</b> | Exploratory Endpoints |
| To explore the effect of once-weekly doses of SYNT001 at different dose levels and dosing durations on biomarkers to understand the pathophysiology of the disease and the SYNT001 mechanisms of action | The exploration of SYNT001 mechanisms of action and effects of SYNT001 on pathophysiology summarized by cohort and timepoint as determined by: Complement component 3 (C3) levels by nephelometry Anti-epithelial cell antibody (AECA) titers by indirect immunofluorescence Fc gamma R2A receptor (FCGR2A) single nucleotide polymorphisms (SNP) by genotyping Presence of disease and inflammatory markers by RNAseq (RNA sequencing) Immunophenotyping via measures of T cells, monocytes, NK cells and B cells by flow cytometry Urine IgG levels to explore SYNT001 distribution and elimination Exploratory biomarkers to investigate immune response associated with pemphigus |

| | To determine the impact of different SYNT001 dose levels and dosing durations on the subject's use of corticosteroids to treat their pemphigus (vulgaris or foliaceus) To assess the impact of once-weekly doses of SYNT001 on the subject's health-related quality of life (HR-QoL) at different dose levels and dosing durations | The evaluation of corticosteroid use during the study will be summarized by cohort and timepoint The assessment of SYNT001 impact on subject's health-related quality of life (HR-QoL) by responses to the Autoimmune Bullous Diseases Quality of Life (ABQoL) questionnaire and Skindex-29 scores summarized by cohort and timepoint |
|---|---|---|
| | To assess the effect of once-weekly doses of SYNT001 on the appearance of skin and mucosal lesions at different dose levels and dosing durations | The qualitative assessment of changes in appearance of skin and mucosal lesions as determined by photography presented by cohort and timepoint |
| | To quantify the amount of SYNT001 in skin (skin biopsies optional) | The determination of SYNT001 levels in skin biopsies across timepoints (skin biopsies optional) |
| Study design | This is a multicenter, open-label safety study to determine the dose regimen of SYNT001 administered intravenously in subjects with pemphigus (vulgaris or foliaceus). Approximately 20 (up to a maximum of 32) eligible subjects with a diagnosis of active pemphigus vulgaris or pemphigus foliaceus will receive planned doses of 10 mg/kg up to 45 mg/kg of SYNT001. Eligible subjects will be enrolled in Cohort 1 and then sequential cohorts, pending recommendation received from the scheduled Dose Escalation Committee (DEC) review. The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organization review the data and participate in the discussions. Each cohort must be fully enrolled before a successive cohort will be opened for enrollment. Cohort 4 is optional and will be added at the discretion of the sponsor and/or DEC. An overview of the study cohorts is provided in Table 1 and Figure 1 shows a schematic of the study design. | |

| Table 1. | <b>Cohort Overview</b> | | | |
|---|---|---|---|---|
| Cohort<br>No. | No. of<br>Subjects | SYNT001<br>Dose | No. of<br>Doses | DEC Review Timepoint |
| 1ª | up to 8 | 10 mg/kg | 5 | NA |
| 2 <sup>b</sup> | 4° | ≤30 mg/kg <sup>d</sup> | 5 | When 100% of Cohort 1 subjects reach Day 42 |
| 3 <sup>b</sup> | 4° | ≤30 mg/kg <sup>d</sup> | 14 | When 50% of Cohort 2 subjects reach Day 42 |
| 4 <sup>b</sup> (optional) | 4 <sup>c</sup> | ≤45 mg/kg <sup>d</sup> | ≤14 | When 50% of Cohort 3 subjects reach Day 42 <sup>e</sup> |

Abbreviations: DEC = Dose Escalation Committee; NA = not applicable

- a. No more than 3 subjects with pemphigus foliaceus may be enrolled
- b. Two or fewer subjects with pemphigus foliaceus may be enrolled
- c. Up to 4 additional subjects may be added following DEC's evaluation.
- d. Dose will be recommended by the DEC and will be based on both an ongoing and set timepoint review of safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities (DLTs), adverse events (AEs), treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and total IgG levels.
- e. All available data will be considered.

The first 2 subjects in Cohorts 1 and 2 will be enrolled at staggered intervals to facilitate adequate safety evaluation before dosing of subsequent subjects may proceed. A staggered dosing interval for the first 2 subjects enrolled in successive cohorts will not be required if the planned dose is equal to or lower than that previously administered.

At 24-hour and 7-day intervals described below, the DEC will review all available safety data (including but not limited to dose limiting toxicities [DLTs], AEs, TEAEs, and SAEs, PD (including but not limited to total IgG levels), and clinical outcomes.

### DEC Safety Review of 24-hour Data for Cohorts 1 and 2, Subject 1

• The first 2 subjects will be dosed at least 24 hours apart. A DEC review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject.

### DEC Safety Review of 7-day Data for Cohorts 1 and 2, Subjects 1 and 2

• The 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining subjects in the cohort.

The 24-hour and 7-day reviews will consider seriousness and severity of AEs/TEAEs/SAEs and relatedness to study drug, vital sign assessments, physical examinations, and clinical laboratory testing.

At scheduled reviews, the DEC may recommend increasing the number of subjects to be enrolled (from 4 up to 8 as shown in Table 1) and advise on the planned dose for each successive cohort. Further, the DEC may recommend pausing and resuming or halting enrollment.

Further, at any time during the study, the DEC may review all available safety data (including but not limited to DLTs, AEs, TEAEs, and SAEs), PD (including but not limited to IgG levels), and clinical outcomes.

- If 2 or more subjects at any time in any cohort have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. Upon review of the available information, the DEC may reduce the dose prior to enrolling additional subjects using the guidelines below:
  - Cohort 1: Dose may be reduced by at least 50%.
  - Cohort 2: Dose may be reduced by at least 33%.
  - Cohort 3: Dose may be reduced to a level lower than the Cohort 2 dose.
  - Cohort 4 (optional cohort): Dose may be reduced to level lower than the Cohort 3 dose.

NOTE: DLT will be defined generally as severe (Grade 3) AEs occurring in ≥2 subjects that are determined to be clinically significant and considered related to study drug.

- If any subject at any time during the study experiences a life-threatening AE (Grade 4) that is related to study drug, further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the appropriate course of action.
- At any time during the study, the study or any ongoing study cohort may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects.

Additional information on the DEC's responsibilities as they pertain to data review, dose selection, opening and closing a cohort, individual and study stopping recommendations is provided in Section 9 and the DEC charter.

### Study methodology

Study participation requires that the subject will have completed the following periods of assessment to be performed on a weekly basis: Screening, Treatment (Baseline [Day 0], Major and Minor Dosing Visit days), and a Follow-Up (Major and Minor Visit days).

Throughout the study, during each period of assessment to evaluate safety and tolerability, subjects will undergo physical examinations (including weight), vital sign measurements (including pulse oximetry), clinical (safety) laboratory tests, AEs, concomitant medication assessments, and ECGs.

### Screening Period (up to 14 days)

After the subject has provided written informed consent, the Investigator or other qualified study personnel will determine if the subject is eligible for the study. This will be accomplished by reviewing the inclusion and exclusion criteria, and the subject's demographic profile, screening PDAI total activity score, and medical history.

Treatment Period (28 or 91 days)

The treatment period includes the Baseline (Day 0) Dosing Visit day, and Major and Minor Dosing Visit days. Refer to Table 2, Table 3, Table 4, and Section 7.

Baseline (Day 0) Visit Day

In addition to the safety and tolerability assessments described above, the subject will be administered the study drug and the following procedures will be conducted: pregnancy test (if applicable), PDAI, PK, PD, and immunogenicity sample collection, photography of lesions, and serum tetanus and varicella zoster virus (VZV) antibody tests. An optional skin biopsy may be collected. HR-QoL is assessed in all cohorts except Cohort 1. A complete list of assessments is provided in Table 2, Table 3, Table 4, and Section 7.

Major Dosing Visit Days

In addition to the safety and tolerability assessments described above, the subject will be administered the study drug, and the following procedures will be conducted: PDAI, PD, and immunogenicity sample collection. A complete list of assessments is provided in Table 2, Table 3, Table 4, and Section 7.

Minor Dosing Visit Days

In addition to the safety and tolerability assessments described above, the subject will be administered the study drug, and the following procedures will be conducted: PDAI and PD sample collection. A complete list of assessments is provided in Table 2, Table 3, Table 4, and Section 7.

### Follow-up Period/End of Study (84 days)

The follow-up period includes the Major and Minor Follow-up Visit days. Subjects are encouraged to participate in all visits up to and including Day 112 (Cohorts 1 and 2) or Day 175 (Cohort 3) to ensure study completion. Refer to Table 2, Table 3, Table 4, and Section 7.

Major Follow-up Visit Days

In addition to the safety and tolerability assessments described above, the following procedures will be conducted: PDAI, PD sample collection, photography of lesions and HR-QoL assessments. A complete list of assessments is provided in Table 2, Table 3, Table 4, and Section 7.

Minor Follow-up Visit Days

In addition to the safety and tolerability assessments described above, the following procedures will be conducted: PDAI and PD sample collection. A complete list of assessments is provided in Table 2, Table 3, Table 4, and Section 7.

Dosing for any individual subject will be discontinued (ie, further treatment with the study drug will not be given) if the subject experiences any study drug-related SAE or any study drug-related non-serious adverse event that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) suggests that it could be unsafe to administer further study drug to that subject. Additionally, a subject will be discontinued from further treatment with study drug at the discretion of the Investigator, with consultation with the Medical Monitor if desired, if they require a significant increase in anti-pemphigus medications for the management of pemphigus.

| Study population | Male or female subjects aged 18 and older with pemphigus (vulgaris or | | |
|---|---|--|--|
| Study population | foliaceus) in active stage | | |
| Inclusion criteria | Subjects must meet the following criteria to be included: | | |
| inclusion criticia | Willing and able to read, understand, and sign an informed consent form. | | |
| | <ol> <li>Withing and able to read, understand, and sign an informed consent form.</li> <li>Male or female ≥18 years of age at the time of screening.</li> </ol> | | |
| | Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 | | |
| | of the following criteria: | | |
| | <ul> <li>a. Documented clinical history consistent with pemphigus vulgaris or<br/>foliaceus (clinical presentation defined as mucosal and/or skin<br/>lesions).</li> </ul> | | |
| | b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal (ULN). | | |
| | c. History of at least one positive tissue-based test (eg, biopsy, direct immunofluorescence [DIF]). | | |
| | 4. Active disease defined as lesions lasting >2 weeks, and 3 active lesions in | | |
| | skin or mucosa or 2 active lesions with at least one being a skin lesion | | |
| | >1 cm diameter: | | |
| | a. If treated with rituximab or other anti-CD20 mAb, last dose >12 months prior to screening. | | |
| | <ul><li>b. If being treated with other immunosuppressants (ie, azathioprine,</li></ul> | | |
| | mycophenolate mofetil, methotrexate, dapsone, cyclosporine, | | |
| | tacrolimus, sirolimus, or low-dose cyclophosphamide | | |
| | [\le 100 mg/day]), dose must be stable, defined as <25% change in | | |
| | dose, for 4 weeks prior to screening. | | |
| | c. On stable dose of corticosteroids, defined as ≤1 mg/kg of | | |
| | prednisone or equivalent and may not be increased by more than | | |
| | 50% in the 2 weeks prior to screening. | | |
| | d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth. | | |
| | e. Stable use of topical low strength hydrocortisone ( $\leq 1\%$ ), | | |
| | tacrolimus, sirolimus, or pimecrolimus for lesions contributing | | |
| | <10% of the PDAI total activity score for the 4 weeks prior to | | |
| | screening is allowed. Stable use of dexamethasone elixir solution | | |
| | (swish and spit only) for oral lesions for the 4 weeks prior to | | |
| | screening is allowed. | | |
| | f. If not on regular corticosteroids, no pulse corticosteroids are allowed in the 2 weeks prior to screening. | | |
| | 5. Body mass index (BMI) >18.5 kg/m <sup>2</sup> . | | |
| | 6. Has a negative pregnancy test documented prior to the first dose of study | | |
| | drug (for women of childbearing potential). | | |
| | 7. Females of childbearing potential must agree to be abstinent or else use | | |
| | any two of the following medically acceptable forms of contraception | | |
| | (<1% per year failure rate) from the screening period through the final | | |
| | study visit: oral contraceptive, condom with or without spermicidal jelly, | | |
| | diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). A female whose male partner has had a vasectomy must agree to | | |
| | use one additional form of medically acceptable contraception. | | |
| <b>r</b> | , |
|---|---|
| | 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or |
| | post-menopausal for at least 12 months do not require contraception |
| | during the study. |
| | 9. Males with female partners of childbearing potential, including males who |
| | are surgically sterile (post vasectomy), must agree to be abstinent or else |
| | use a medically acceptable form of contraception from the screening |
| | period through 60 days after the final study visit. |
| 7 | 10. A PDAI total activity score of >4 at screening. |
| Exclusion criteria | Subjects meeting any of the following criteria are to be excluded: |
| | 1. Subject unable or unwilling to comply with the protocol. |
| | 2. Active non-hematologic malignancy or history of non-hematologic |
| | malignancy in the 3 years prior to screening (exclusive of non-melanoma |
| | skin cancer and cervical cancer in situ). 3. Positive for human immunodeficiency virus (HIV) or hepatitis C antibody. |
| | 4. Positive for hepatitis B surface antigen. |
| | 5. Active infection or history of recurrent infections. |
| | 6. IVIG treatment within 30 days of screening. |
| | 7. Received any cytotoxic (other than azathioprine) or any non-anti-CD20 |
| | mAb therapy in the 3 months prior to screening. |
| | 8. Any exposure to an investigational drug or device within the 30 days prior to screening. |
| | 9. Plasmapheresis or immunoadsorption within 30 days of screening. |
| | 10. Cellular therapy, including chimeric antigen receptor and T-cell (CAR-T), at any time prior to screening. |
| | 11. Use of any systemic or topical immunosuppressive drugs within 3 months |
| | of screening not including dose allowed by the inclusion criteria. |
| | 12. Serum total IgG <600 mg/dL. |
| | 13. Subject has any current medical condition that, in the opinion of the |
| | Investigator, may compromise their safety or compliance, preclude |
| | successful conduct of the study, or interfere with interpretation of the results (eg, a significant pre-existing illness or other major comorbidity |
| | that the Investigator considers may confound the interpretation of the |
| | study results). |
| | 14. Any vaccination within 2 weeks of screening. |
| Study drug, dosage, | Study drug: SYNT001 |
| and administration | Dosage: |
| | Cohort 1: 10 mg/kg, 5 weekly IV doses |
| | Cohort 2: ≤30 mg/kg, 5 weekly IV doses |
| | Cohort 3: ≤30 mg/kg, 14 weekly IV doses |
| | Cohort 4 (optional cohort): ≤45 mg/kg, ≤14 weekly IV doses |
| | Product presentation and preparation: |
| | SYNT001 provided as a liquid at a nominal concentration of 50 mg/mL. SYNT001 is diluted in dextrose 5% in water (D5W) to prepare the solution for infusion. |
| | Route of administration: IV in 250 mL over 1 hour ± 15 minutes |
| | Noute of authinistration: 1 v III 250 IIIL over 1 hour ± 15 minutes |

| Control, dose, and | Not applical | ole | | | | |
|---|---|---|---|---|---|---|
| route of administration | | | | | | |
| Duration of subject | The duration | n of subject no | articipation fo | r each cohort | is as follow | c· |
| participation | Cohorta | Screening | Treatment | Follow-up | Maximum | |
| | Conort | Sercening | Treatment | 1 onow up | Days | Weeks |
| | 1 | ≤14 days | 28 days | 84 days | 126 days | 18 weeks |
| | 2 | ≤14 days | 28 days | 84 days | 126 days | 18 weeks |
| | 3 | ≤14 days | 91 days | 84 days | 189 days | 27 weeks |
| | | | | • | , | al cohort) will be |
| | | | EC data review. | | | |
| Permitted and | | • | eceives within | • • | or to enrollm | ent through |
| prohibited | | - | e documented | d. | | |
| concomitant<br>treatments | | Medications | | | | |
| treatments | | | and treatment | | _ | s, including |
| | 1 | | permitted if no | - | | |
| | | | treat active in | | | g the study. |
| | _ | 2. Topical or systemic treatments for oral candidiasis. | | | | |
| | | <ul><li>3. Topical lidocaine for transient pain relief as needed.</li><li>4. Concomitant treatment that is medically indicated for any AEs the subject</li></ul> | | | | |
| | | experiences during the study. | | | | |
| | 5. Medicat | ion for potent | ial infusion re | eactions: The | Investigator | may |
| | | | ctic use of ace | | | |
| | - | • | , , | . • | ranitidine, fa | amotidine), etc |
| | | | nfusion reaction | | e <1%) annli | ed to a single |
| | | | .0% of the PD | | | ed to a single |
| | 7. Topical | tacrolimus, si | rolimus or pir<br>the PDAI total | mecrolimus a | pplied to a s | ingle lesion |
| | | - | solution for o | • | | ıs stable |
| | | | ipation (swisl | | | 15 544615 |
| | | | following sys | | | |
| | | | | | | , cyclosporine, |
| | | | | | | (100 mg/day). |
| | | | on. <b>Prohibite</b> | | | be tapered at |
| | | | | | | e study unless |
| | | ove as permit | | iot de perimi | ica during in | e study unless |
| | | | ti-CD20 antil | • | | |
| | | | es other than s | | | |
| | | ical or system<br>d as permitted | ic immunosu | ppressive dru | igs apart froi | n those that |
| | | - | or to infusion | (except in su | biects who r | eceived |
| | | | atment of a pr | | | |
| | | tary herbal su | | | 2 | <del>-</del> / |
| | 6. Any inv | estigational d | rug or device | | | |
| | | | weeks of scr | eening throu | gh 28 days fo | ollowing final |
| | dose of | study drug | | | | |

# Statistical considerations

Three populations will be employed in the analysis of study data:

- The safety population will consist of all subjects who have received at least one dose of study drug.
- The PD population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.
- The PK population will consist of all subjects who receive at least one dose of study drug and have post-dose PK data available.

Primary safety analyses will be performed on the safety population. Demographics, subject disposition, screening, and baseline characteristics will be summarized for the safety and PD/PK populations, where appropriate.

#### Sample size

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

#### Criteria for evaluation

Baseline analysis

Baseline characteristics to include medical history, physical examination, vital signs, and ECG will be summarized using descriptive statistics by cohort.

#### Safety analysis

The evaluation of SYNT001 based on vital signs, physical examination, ECGs, clinical safety laboratory tests, the incidence of AEs, TEAEs, and SAEs summarized by cohort, severity, and relationship to study product.

#### Dose-finding analysis

The evaluation of SYNT001 based on total IgG levels and responses on the PDAI total activity score from baseline will be summarized using descriptive statistics by cohort.

#### Statistical methodology

Treatment-emergent AEs (TEAEs) will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least one occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject and dose using SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by time point and cohort. The incidence of laboratory abnormalities will be summarized. The worst on-study grade

after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, or above the normal limits of the central laboratory. Vital sign measurements will be summarized by cohort at each scheduled time point using descriptive statistics. PD/PK results will be summarized by cohort. Descriptive statistics of PD/PK parameters for SYNT001 will include mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum Immunogenicity results will be summarized by cohort and timepoint. Descriptive statistics will include mean, SD, median, minimum, and maximum.

PDAI results will be summarized by score (total activity score, total damage score), cohort, and timepoint. Descriptive statistics will include absolute change from baseline and percent change from baseline.

Figure 1. Cohort Enrollment



**Table 2.** Study Assessments for Cohort 1

| | Screening | | | | | | | Tre | atment | Period | | | | | | | Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 |
| Time point (study day) | -14 to -1 | 0 | 1 | 2 | 5 <sup>p</sup> | 7 | 12 <sup>p</sup> | 14 | 19 <sup>p</sup> | 21 | 28 | 29 | 30 | 33 | 42 | 56 | 84 | 112 or |
| | | | (±1 h) | (±2 h) | (±4 h) | (±6 h) | (±6 h) | (±6 h) | (±6 h) | (±6 h) | (±6 h) | (±1 h) | (±2 h) | (±4 h) | (±3 d) | (±5 d) | (±5 d) | ET (±5 d) |
| Informed consent | X | | | | | | | | | | | | | | | | | |
| Demographics/medical history | X | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | | | | | | | | |
| Physical examination <sup>a</sup> | X | X | | | | X | | X | | X | X | | | | X | X | X | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>c</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Clinical safety labs <sup>d</sup> | X | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis and HIV screen | X | | | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>f</sup> | X | X | | | | | X | | | | X | | | | | X | | |
| Tetanus and VZV antibodies <sup>g</sup> | | X | | | | | | | | | | | | | | X | X | X |
| PDAI | | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| PK sampling <sup>h</sup> | | X | X | X | X | | | | | | X | X | X | X | | | | |
| Immunogenicity <sup>i</sup> | | X | | | | | | X | | | X | | | | | X | X | X |
| Study drug administration <sup>j</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4) <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Xq |
| CIC | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Anti-Dsg (1 and 3) antibody titers | X | X | | | | X | | X | | | | | | X | | X | X | X |
| C3 and AECA <sup>1</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| FCGR2A by buccal swab <sup>m</sup> | | X | | | | | | | | | | | | | | | | |
| RNAseq | | X | | | | | | X | | | | | | X | | X | X | X |
| Urine IgG | | X | | | | | | X | | | | | | X | | X | X | X |
| Immunophenotyping <sup>n</sup> | | X | | | | | | | | | X | | | | | X | | |
| Exploratory pemphigus immune response biomarkers | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Optional skin biopsy | | X | X | X | | | | X | | | | | | X | | X | X | |
| Photography <sup>o</sup> | | X | | | | | | | | | | | | X | | X | X | X |
| Adverse events | | | | | To be c | ollected | from the | e date th | at the IC | CF is sig | ned thro | ugh the | last stud | ly visit | | | | |
| Concomitant medications | | | | | | | from wi | | | | | | | | | | | |

Abbreviations: CIC = circulating immune complexes; d = days; ECG = electrocardiogram; ET = early termination; h = hour(s); HIV = human immunodeficiency virus; ICF = informed consent form; PDAI = Pemphigus Disease Area Index; PK = pharmacokinetic; VZV = varicella zoster virus.

- a. Complete physical examination, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.
- b. **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. On Days 0, 7, 14, 21, and 28, vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour, and 2 hours following completion of the infusion.
- c. **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d. Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 7.5 for a complete list). Full clinical safety laboratory draws will be collected at screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84, and 112.
- e. **Pregnancy test**: To be performed at time of screening, prior to first dose of SYNT001 on Day 0, and on Days 56 and 112. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.
- f. Digital 12-lead ECG to be obtained in triplicate at least 1 to 2 minutes apart and after 5 minutes of rest in a supine position. See Section 7.6 for additional information. On Days 0 and 28 to be obtained 5 minutes after the completion of infusion. Day 12 ECG will be collected only if the visit is conducted at the study site.
- g. **Serology**: Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 84; if still below the baseline value (or level of detection), the subject will be re-tested at Day 112. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112, will be referred to their primary care physician for further management. See Section 7.5.3 for additional information.
- h. **PK**: Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. See Section 7.5.4 for additional information.
- i. Immunogenicity: Samples will be collected pre-dose when collected on dosing days. Samples will be collected on Days 0, 14, 28, 56, 84 and 112. See Section 7.5.6 for additional information.
- j. Prior to **study drug infusion**, SYNT001 drug product is to be diluted in dextrose 5% in water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour using a 0.2-micron inline filter. See Section 4 and Section 7.8 for additional information.
- k. Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 7.5.5 for additional information.
- 1. **Exploratory pharmacodynamic samples (C3 and AECA):** Collected pre-dose when collected on dosing days. See Section 7.5.5 for complete information.
- m. Buccal samples to be collected and stored; pending review of clinical and pharmacodynamics assessments.
- n. Immunophenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells.
- o. Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- p. Visit Days 5, 12, and 19 may be conducted via at-home nurse in lieu of a subject visit to the study site.
- q. Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

Table 3. Study Assessments for Cohort 2

| | Screening | | Tr | eatment Per | iod | | | | Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 |
| Time point (study day) | -14 to -1 | 0 | 7<br>(±1 d) | 14<br>(±1 d) | 21<br>(±1 d) | 28<br>(±1 d) | 35<br>(±1 d) | 42<br>(±1 d) | 56<br>(±3 d) | 84<br>(±5 d) | 112 or ET (±5 d) |
| Informed consent | X | | | | | | | | | | |
| Demographics/medical history | X | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | |
| Physical examination <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>c</sup> | | X | X | X | X | X | | | | | |
| Clinical safety labs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | X | | X |
| Hepatitis and HIV screen | X | | | | | | | | | | |
| 12-lead ECG <sup>f</sup> | X | X | | X | | X | | | X | | |
| Tetanus and VZV antibodies <sup>g</sup> | | X | | | | | | | X | | X |
| PDAI <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X |
| PK sampling <sup>i</sup> | | X | | | | X | | | | | |
| Immunogenicity <sup>j</sup> | | X | | X | | X | | | X | | X |
| Study drug administration <sup>k</sup> | | X | X | X | X | X | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4) <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | $X^q$ |
| CIC | | X | X | X | X | X | X | X | X | X | X |
| Anti-Dsg (1 and 3) antibody titers | X | X | X | X | X | X | X | X | X | X | X |
| C3 and AECA <sup>m</sup> | | X | | | | | X | | X | | |
| FCGR2A by buccal swab <sup>n</sup> | | X | | | | | | | | | |
| RNAseq | | X | | | | | X | | X | | |
| Urine IgG | | X | | | | | X | | X | | |
| Immunophenotyping <sup>o</sup> | | X | | | | | X | | X | | |
| Exploratory pemphigus immune response biomarkers | | X | X | X | X | X | X | X | X | X | X |
| Photography <sup>p</sup> | | X<br>X | | | | | X | | X | | X |
| HR-QoL assessments | | X | | | | | X | | X | | X |
| Adverse events | | - | To be | collected from | n the date the | at the ICF is s | igned throug | h the last stu | dy visit | | |
| Concomitant medications | | | To be | collected from | n within 14 a | lays prior to l | Day 0 through | h th <mark>e last stud</mark> | ly visit | | |

Abbreviations: CIC = circulating immune complexes; d = day(s); ECG = electrocardiogram; ET = early termination; HIV = human immunodeficiency virus; HR-QoL = health-related quality of life; ICF = informed consent form; PDAI = Pemphigus Disease Area Index; PK = pharmacokinetic; VZV = varicella zoster virus.

a. Complete physical examination, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.

b. **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. Vital sign measurements will be taken on all study visits. On Days 0, 7, 14, 21, and 28, vital sign measurements

- will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour, and 2 hours following completion of the infusion.
- c. **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d. Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 7.5 for a complete list). Full clinical safety laboratory draws will be collected at screening and on all study visits.
- e. **Pregnancy test**: To be performed at time of screening, prior to first dose of SYNT001 on Day 0, and on Days 56 and 112. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.
- f. Digital 12-lead ECG to be obtained in triplicate at least 1 to 2 minutes apart and after 5 minutes of rest in a supine position. See Section 7.6 for additional information. On treatment days to be obtained 5 minutes after the completion of infusion.
- g. **Serology**: Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline and is not within 30% of the baseline value or is below the protective level by End of Treatment will be referred to their primary care physician for further management. See Section 7.5.3 for additional information.
- h. **PDAI** will be administered at screening. Subject eligibility requires a PDAI total activity score >4. Thereafter, assuming eligibility, the PDAI will be administered during Treatment Period and Follow-up Period. See Section 7.7 for additional information.
- i. **PK**: On Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes, 1 and 2 hours after the end of study drug infusion. See Section 7.5.4 for additional information.
- j. **Immunogenicity**: Samples will be collected pre-dose when collected on dosing days. Samples will be collected on Days 0, 14, 28, 56, and 112. See Section 7.5.6 for additional information.
- k. Prior to **study drug infusion**, SYNT001 drug product is to be diluted in dextrose 5% in water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour ± 15 minutes using a 0.2-micron inline filter. See Section 4 and Section 7.8 for additional information.
- 1. **Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4):** Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 7.5.5 for additional information.
- m. Exploratory pharmacodynamic samples (C3 and AECA): Collected pre-dose when collected on dosing days. See Section 7.5.5 for complete information.
- n. Buccal samples to be collected and stored; pending review of clinical and pharmacodynamics assessments.
- o. Immunophenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells.
- p. Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 35, 56, and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- q. Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

Table 4.Study Assessments for Cohort 3

| | Screening | | | | | | , | Treatm | ent Per | iod | | | | | | | F | ollow-U | <sup>J</sup> p | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| Time point (study day) | -14 to -1 | 0 | 7<br>(±1 d) | 14<br>(±1 d) | 21<br>(±1 d) | 28<br>(±1 d) | 35<br>(±1 d) | 42<br>(±1 d) | 49<br>(±1 d) | 56<br>(±1 d) | 63<br>(±1 d) | 70<br>(±1 d) | 77<br>(±1 d) | 84<br>(±1 d) | 91<br>(±1 d) | 98<br>(±1 d) | 105<br>(±1 d) | 119<br>(±3 d) | 147<br>(±5 d) | 175 or<br>ET<br>(±5 d) |
| Informed consent | X | | | | | | | | | | | | | | | | | | | |
| Demographics/medical history | X | | | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | | | | | | | | | | |
| Physical examination <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>c</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | |
| Clinical safety labs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | | | | X | | | | | | | X | | | X | | X |
| Hepatitis and HIV screen | X | | | | | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>f</sup> | X | X | | | | | | X | | | | | | | X | | | X | | |
| Tetanus and VZV antibodies <sup>g</sup> | | X | | | | | | | | | | | | | | | | X | | X |
| PDAI <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PK sampling <sup>i</sup> | | X | | | | | | | | | | | | | X | | | | | |
| Immunogenicity <sup>j</sup> | | X | | | | | | X | | | | | | | X | | | X | | X |
| Study drug administrationk | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | | | | |
| Immunoglobulins <sup>l</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | $X^q$ |
| CIC | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Anti-Dsg (1 and 3) antibody titers | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| C3 and AECA <sup>m</sup> | | X | | | | | | | | | | | | | | X | | X | | |
| FCGR2A by buccal swab <sup>n</sup> | | X | | | | | | | | | | | | | | | | | | |
| RNAseq | | X | | | | | | | | | | | | | | X | | X | | |
| Urine IgG | | X | | | | | | | | | | | | | | X | | X | | |
| Immunophenotyping <sup>o</sup> | | X | | | | | | | | | | | | | | X | | X | | |
| Exploratory pemphigus immune response biomarkers | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Photography <sup>p</sup> | | X | | | | | | X | | | | | | | | X | | X | | X |
| HR-QoL assessments | | X | | | | | | | | | | | | | | X | | X | | X |
| Adverse events | | | | | 7 | o be co | llected t | rom the | date th | at the IC | CF is sig | ned thr | ough the | e last sti | udy visit | | | | | |
| Concomitant medications | | | | | | | | | | | | | | | ıdy visit | | | | | |

Abbreviations: CIC = circulating immune complexes; d = days; ECG = electrocardiogram; ET = early termination; HIV = human immunodeficiency virus; ICF = informed consent form; PDAI = Pemphigus Disease Area Index; PK = pharmacokinetic; VZV = varicella zoster virus.

a. Complete physical examination, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.

b. Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. Vital sign measurements will be taken on all study visits. On Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84,

- and 91, vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour, and 2 hours following completion of the infusion.
- c. **Pulse oximetry:** On Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, and 91, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d. Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 7.5 for a complete list). Full clinical safety laboratory draws will be collected at screening and on all study visits.
- e. **Pregnancy test**: To be performed at time of screening, prior to dosing of SYNT001 on Days 0, 42, and 91, and on Days 119 and 175. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.
- f. Digital 12-lead ECG to be obtained in triplicate at least 1 to 2 minutes apart and after 5 minutes of rest in a supine position. See Section 7.6 for additional information. On treatment days to be obtained 5 minutes after the completion of infusion.
- g. **Serology**: Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the protective level by End of Treatment will be referred to their primary care physician for further management. See Section 7.5.3 for additional information.
- h. **PDAI** will be administered at screening. Subject eligibility requires a PDAI total activity score >4. Thereafter, assuming eligibility, the PDAI will be administered during Treatment Period and Follow-up Period. See Section 7.7 for additional information.
- i. **PK**: Starting on Days 0 and 91, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes, 1 hour and 2 hours after the end of study drug infusion. Section 7.5.4 for additional information.
- j. Immunogenicity: Samples will be collected pre-dose when collected on dosing days. Samples will be collected on Days 0, 42, 91, 119 and 175. See Section 7.5.6 for additional information.
- k. Prior to **study drug infusion**, SYNT001 drug product is to be diluted in dextrose 5% in water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour ± 15 minutes using a 0.2-micron inline filter. See Section 4 and Section 7.8 for additional information.
- 1. **Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4):** Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, IgM at every visit. On Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, and 91, samples are collected prior to infusion of study drug. See Section 7.5.5 for additional information.
- m. Exploratory pharmacodynamic samples (C3 and AECA): Collected pre-dose when collected on dosing days. See Section 7.5.5 for complete information.
- n. Buccal samples to be collected and stored; pending review of clinical and pharmacodynamics assessments.
- o. Immunophenotyping by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, NK cells and B cells.
- p. Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 42, 98, 119, and 175. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- q. Subjects will return to the clinic on Days 147 and 175 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 175 visit will be referred for further management.

## TABLE OF CONTENTS

| 1. | SYN | NOPSIS | 4 |
|-----|-------|----------------------------------|----|
| LIS | ST OF | TABLES | 27 |
| LIS | ST OF | FIGURES | 27 |
| LIS | ST OF | APPENDICES | 27 |
| LIS | ST OF | ABBREVIATIONS | 28 |
| 2. | BAG | CKGROUND AND RATIONALE | 31 |
| | 2.1 | Study Rationale | 31 |
| | 2.2 | Selection of Doses in this Study | 32 |
| | 2.3 | Compliance Statement | 33 |
| 3. | STU | JDY OBJECTIVES AND ENDPOINTS | 34 |
| | 3.1 | Primary Objective | 34 |
| | 3.2 | Secondary Objectives. | 34 |
| | 3.3 | Exploratory Objectives | 34 |
| | 3.4 | Primary Endpoints | 34 |
| | 3.5 | Secondary Endpoints | 35 |
| | 3.6 | Exploratory Endpoints | 35 |
| 4. | STU | JDY DRUG | 37 |
| | 4.1 | Description of SYNT001 | 37 |
| | 4.2 | Dose Requirements | 37 |
| | 4.3 | Handling and Storage of SYNT001 | 37 |
| | 4.4 | Study Drug Accountability | 37 |
| 5. | STU | JDY DESIGN | 39 |
| | 5.1 | Study Sites | 39 |
| | 5.2 | Overview of Study Design | 39 |
| | 5.3 | Randomization and Blinding | 40 |
| 6. | STU | JDY POPULATION | 41 |
| | 6.1 | Target Population | 41 |
| | 6.2 | Inclusion Criteria | 41 |
| | 6.3 | Exclusion Criteria | 42 |
| 7. | STU | JDY PROCEDURES | 44 |
| | 7.1 | Informed Consent | 44 |
| | 7.2 | Demographics and Medical History | 44 |
| | 7.3 | Physical Examination. | 44 |
| | 7.4 | Vital Sign Measurements | 44 |
| | 7.5 | Clinical Laboratory Measurements | 46 |
| | 7 | .5.1 Pregnancy Testing | 47 |
| | 7 | .5.2 Virology | 47 |

| | 7.5 | 5.3 | Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing47 | 7 |
|---|---|---|---|---|
| | 7.5 | 5.4 | Pharmacokinetics (PK) Sampling | 7 |
| | 7.5 | 5.5 | Pharmacodynamic Sampling47 | 7 |
| | 7.5 | 5.6 | Immunogenicity Testing | 3 |
| | 7.6 | 12-L | ead Electrocardiogram (ECG)49 | 9 |
| | 7.7 | Pemp | phigus Disease Area Index (PDAI) | 9 |
| | 7.8 | Study | y Drug Administration | 9 |
| | 7.9 | Photo | ographs49 | 9 |
| | 7.10 | Healt | th-Related Quality of Life Assessments50 | ) |
| | 7.11 | Adve | erse Event Assessments | ) |
| | 7.12 | Prior | and Concomitant Medications | ) |
| | 7.13 | Skin | Biopsy5 | 1 |
| 8. | STU | DY AS | SSESSMENTS52 | 2 |
| | 8.1 | All C | Cohorts: Screening Period and First Treatment (Day 0) | 2 |
| | 8.1 | 1.1 | All Cohorts: Screening Period (Day -14 to Day -1)52 | 2 |
| | 8.1 | 1.2 | All Cohorts: Enrollment and First Treatment (Day 0) | 2 |
| | 8.2 | Coho | ort 1: Day 1 to 8454 | 4 |
| | 8.2 | 2.1 | Cohort 1: Follow-up Day 1 | 4 |
| | 8.2 | 2.2 | Cohort 1: Follow-up Day 2 | 4 |
| | 8.2 | 2.3 | Cohort 1: Follow-up Day 554 | 4 |
| | 8.2 | 2.4 | Cohort 1: Treatment Day 7 (Dose 2)55 | |
| | 8.2 | 2.5 | Cohort 1: Follow-up Day 1255 | 5 |
| | 8.2 | 2.6 | Cohort 1: Treatment Day 14 (Dose 3) | |
| | 8.2 | 2.7 | Cohort 1: Follow-up Day 19 | 7 |
| | 8.2 | 2.8 | Cohort 1: Treatment Day 21 (Dose 4) | |
| | 8.2 | 2.9 | Cohort 1: Treatment Day 28 (Dose 5) | |
| | 8.2 | 2.10 | Cohort 1: Follow-up Day 29 | ) |
| | | 2.11 | Cohort 1: Follow-up Day 30 | |
| | | 2.12 | Cohort 1: Follow-up Day 33 | |
| | | 2.13 | Cohort 1: Follow-up Day 42 | |
| | | 2.14 | Cohort 1: Follow-up Day 5660 | |
| | | 2.15 | Cohort 1: Follow-up Day 84 | |
| | 8.3 | | orts 2 and 3: Subsequent Treatments to Follow-up | 1 |
| | 8.3 | 3.1 | Cohort 2: Treatment Days 7 and 21; Cohort 3: Treatment Days 7, 14, 21, | 1 |
| | 0.0 | , , | 28, 35, 49, 56, 63, 70, 77, and 84 | |
| | | 3.2 | Cohort 2: Treatment Days 14 and 28; Cohort 3: Treatment Days 42 and 916 | |
| | | 3.3 | Cohort 2: Follow-up Days 35 and 56; Cohort 3: Follow-up Days 98 and 119 | 103 |
| | 8.3 | 3.4 | Cohort 2: Follow-up Days 42 and 84; Cohort 3: Follow-up Days 105 and 147 | 4 |
| | | | ± 1 / ·································· | |

| 8.4 | | Cohorts: End of Study or Early Termination Visit; Cohorts 1 and 2 ort 3, Day 175 | • |
|---|---|---|---|
| 9. STU | | ULES | |
| 9.1 | | ect Withdrawal | |
| 9.2 | • | ect Replacement | |
| 9.3 | | ly Discontinuation | |
| 9.4 | | to Follow-up | |
| 9.5 | | ping Rules | |
| 9 | 0.5.1 | Dose-Escalation Stopping Rule | |
| 9 | .5.2 | Study Stopping Rule | |
| 9 | .5.3 | Individual Stopping Rule | |
| 10. EV. | ALUA | ΓΙΟΝ OF SAFETY | |
| 10.1 | Safe | ty Parameters | 69 |
| 10.2 | Adv | erse Events | 69 |
| 1 | 0.2.1 | Recording an Adverse Event | 70 |
| 1 | 0.2.2 | Assessment of Causality | 70 |
| 1 | 0.2.3 | Serious Adverse Events | 70 |
| | 10.2 | .3.1 Recording a Serious Adverse Event | 71 |
| | 10.2 | .3.2 Reporting a Serious Adverse Event | 72 |
| 1 | 0.2.4 | Follow-Up of Adverse Events and Serious Adverse Events | 73 |
| 10.3 | War | nings and Precautions | 73 |
| 1 | 0.3.1 | Vaccinations | 73 |
| 1 | 0.3.2 | Management of Allergic or Infusion-Related Reactions | 73 |
| 1 | 0.3.3 | Potential Immune Effects | 77 |
| 10.4 | Ever | nts of Special Interest | 78 |
| 10.5 | Othe | er Safety Considerations | 78 |
| 1 | 0.5.1 | Laboratory Data | 78 |
| 1 | 0.5.2 | Medication Errors | 79 |
| 1 | 0.5.3 | Overdose | 79 |
| 1 | 0.5.4 | Pregnancy | 79 |
| 11. STA | ATISTI | CAL CONSIDERATIONS | 80 |
| 11.1 | Gene | eral Design | 80 |
| 11.2 | Stud | y Populations | 80 |
| 11.3 | Sam | ple Size Justification | 80 |
| 11.4 | Stati | stical Analysis | 80 |
| 1 | 1.4.1 | Statistical Analysis Plan | 80 |
| 1 | 1.4.2 | Statistical Methodology | 81 |
| 1 | 1.4.3 | Analysis of Primary Endpoints | 81 |

| | 11.4.3 | 3.1 Safety Data | 81 |
|---|---|---|---|
| | 11.4.3 | 3.2 Dose Selection Data | 82 |
| 1 | 1.4.4 | Analysis of Secondary Endpoints | 82 |
| | 11.4.4 | 1.1 Pharmacokinetic Data | 82 |
| | 11.4.4 | 1.2 Pharmacodynamic/Activity Data | 82 |
| | 11.4.4 | Immunogenicity Data | 82 |
| | 11.4.4 | I.4 PDAI Data | 83 |
| 1 | 1.4.5 | Analysis of Exploratory Endpoints | 83 |
| | 11.4.5 | 5.1 Corticosteroid Use | 83 |
| | 11.4.5 | 5.2 Health-Related Quality of Life Data | 83 |
| | 11.4.5 | 5.3 Photography | 83 |
| 11.5 | Interi | m Analysis | 83 |
| 12. STU | DY MA | ANAGEMENT | 84 |
| 12.1 | Regul | atory and Ethical Considerations | 84 |
| 12 | 2.1.1 | Ethical Conduct | 84 |
| 12 | 2.1.2 | Informed Consent | 84 |
| 12 | 2.1.3 | Subject Confidentiality and Privacy | 84 |
| 12 | 2.1.4 | Future Use of Stored Specimens | 85 |
| 12.2 | Study | Administration | 85 |
| 12 | 2.2.1 | Institutional Review Board Approval | 86 |
| 12 | 2.2.2 | Data Handling and Record Keeping | 86 |
| 12 | 2.2.3 | Data Protection | 86 |
| 12 | 2.2.4 | Study Site Regulatory Documentation | 86 |
| 12 | 2.2.5 | Subject Clinical Source Documents and Background Data | 87 |
| 12 | 2.2.6 | Electronic Case Report Forms | 88 |
| 12.3 | Clinic | eal Monitoring, Audits, and Inspections | |
| 12 | 2.3.1 | Clinical Monitoring. | 88 |
| 12 | 2.3.2 | Audits and Inspections | |
| 12.4 | Chang | ges to the Protocol | 89 |
| 12.5 | Study | Discontinuation and Closure | 89 |
| 13. PUE | BLICAT | TON AND DATA SHARING POLICY | 90 |
| 14 REE | FRENC | 252 | 91 |

## LIST OF TABLES

| Table 1.Cohort Overview | 8 |
|---|---|
| Table 2.Study Assessments for Cohort 1 | 17 |
| Table 3.Study Assessments for Cohort 2 | 19 |
| Table 4.Study Assessments for Cohort 3 | 21 |
| Table 5.Cohort Overview | 39 |
| Table 6.Timing Windows for PK/PD Sampling, ECG, and Vital Sign Measurements | 45 |
| Table 7.Clinical Safety Laboratory Panels | 46 |
| Table 8.Pharmacodynamic Assessments | 48 |
| Table 9.Grading and Management of Allergic or Infusion-Related Reactions | 77 |
| Table 10.Study Administrative Structure | 86 |
| LIST OF FIGURES Figure 1.Cohort Enrollment | 16 |
| Figure 2.Management of Moderate (Grade 2) Infusion Reactions | |
| Figure 3.Management of Severe (Grade 3 or Higher) Infusion Reactions | |
| LIST OF APPENDICES | |
| APPENDIX 1.NCI CTCAE, Version 4.03 | 93 |
| APPENDIX 2.Pemphigus Disease Area Index (PDAI) | 174 |
| APPENDIX 3. Autoimmune Bullous Disease Quality of Life (ABQoL) Questionnaire | 175 |
| APPENDIX 4.Skindex-29 | 179 |

#### LIST OF ABBREVIATIONS

Autoimmune Bullous Disease Quality of Life **ABOoL** 

ADA anti-drug antibodies AΕ adverse event

**AECA** Anti-epithelial cell antibody ALT alanine aminotransferase AST aspartate aminotransferase

 $AUC_{0-24}$ area under the plasma concentration-time curve from pre-dose (time<sub>0</sub>) to 24 hours

 $AUC_{0-\infty}$ area under the plasma concentration-time curve from pre-dose (time<sub>0</sub>) to infinity

**BLQ** below the limit of quantification

BMI body mass index BUN blood urea nitrogen

complement component 1q C1q C3 complement component 3

CAR-T chimeric antigen receptor and T-cell

**CFR** Code of Federal Regulations CIC circulating immune complexes

 $C_{\text{max}}$ maximum plasma concentration determined directly from the concentration-time

profile

**CRO** contract research organization

CVcoefficient of variation

**CVID** common variable immune deficiency

D5W dextrose 5% in water

**DEC** Dose Escalation Committee direct immunofluorescence DIF DLT dose-limiting toxicity DNA deoxyribonucleic acid

desmoglein Dsg

**ECG** electrocardiogram

eCRF electronic case report form **EDC** electronic data capture ET early termination

FCGR2A Fc gamma R2a receptor FcRn neonatal Fc receptor

**FDA** Food and Drug Administration

GCP Good Clinical Practice

 $H_2$ histamine<sub>2</sub> **HBV** hepatitis B virus **HCV** hepatitis C virus HIPAA Health Insurance Portability and Accountability Act

HIV human immunodeficiency virus
HR-QoL health-related quality of life
IB Investigator's Brochure
IC immune complex

IC immune complex
ICF Informed Consent Form

ICH International Council on Harmonisation

IgA immunoglobulin A
IgG immunoglobulin G
IgG1-4 immunoglobulin G1-G4
IgM immunoglobulin M
IND investigational new drug
IRB institutional review board

IUD intrauterine IV intravenous

IVIG intravenous immunoglobulin

mAb monoclonal antibody
MED minimum effective dose

MedDRA Medical Dictionary for Regulatory Activities

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NHP nonhuman primate

NOAEL no observed adverse effect level

PD pharmacodynamics

PDAI Pemphigus Disease Area Index

PK pharmacokinetic

QTcF corrected QT interval using Fridericia's formula

RNAseq RNA sequencing
SAE serious adverse event
SAP statistical analysis plan
SAS Statistical Analysis System

SD standard deviation

SNP single nucleotide polymorphism

SOC system organ class

SYNT001 a humanized, affinity matured IgG4-kappa monoclonal antibody

 $t_{1/2}$  Half-life

TEAE treatment-emergent adverse event

T<sub>max</sub> observed time to reach peak plasma concentration

ULN upper limit of normal
US United States of America
VZV varicella zoster virus

WAIHA warm autoimmune hemolytic anemia

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

#### 2. BACKGROUND AND RATIONALE

SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks immunoglobulin G (IgG) and circulating IgG immune complex (CIC) interactions with the neonatal crystallizable fragment receptor (FcRn), and inhibits the varied roles played by FcRn in the immune response.

Through specific and high affinity blockade of FcRn, SYNT001 has been shown to increase the catabolism of IgG and CIC in healthy volunteers and is predicted to block the ability of CIC to activate intracellular signaling events associated with binding to FcRn. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with CICs further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric CIC interactions with FcRn within antigenpresenting cells should result in inhibition of CIC inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of CICs within and among compartments important in cellular immunity, it is further anticipated that SYNT001 will block antigen processing and presentation of antigens contained within CIC that otherwise lead to CD8<sup>+</sup> and CD4<sup>+</sup> T cell activation. Thus, SYNT001 is expected to specifically target immune functions associated with IgG and CIC that are involved in certain IgG-mediated autoimmune conditions.

SYNT001 targets key mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders, including warm autoimmune hemolytic anemia (WAIHA) pemphigus, pemphigoid, myasthenia gravis, immune thrombocytopenic purpura (ITP), and chronic inflammatory demyelinating polyneuropathy (CIDP).

While current treatments for certain autoimmune disorders, including chronic steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 mAbs, such as rituximab, can be effective, they are associated with significant adverse effects, and delayed or non-durable responses.

Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies are thought to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001, which significantly decreases total IgG levels, including a predicted corresponding decrease in the levels of the pathogenic autoantibodies, may lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce CICs and the associated innate and adaptive immune responses may allow for further sustained disease modification.

### 2.1 Study Rationale

This study is being conducted to evaluate the safety, dose, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers.

#### 2.2 **Selection of Doses in this Study**

The SYNT001 dose levels for study SYNT001-103 were selected following careful review of the safety, tolerability, and PD effect on total IgG levels studied in non-human primates (NHP) and healthy male subjects.

8 June 2018

Four repeat-dose toxicology studies in cynomolgus monkeys examined 2 to 14 repeat weekly IV doses 5 to 100 mg/kg SYNT001 with up to a 4-week follow-up. There was one death in the 14week study attributed to an immune-evoked infusion reaction, which correlated with the development of ADAs, circulating immune complexes, circulating complement depletion, and deposition of immune complexes containing SYTN001 and complement in tissues. Across studies, clinical signs were limited to reports of transient emesis/vomitus following dosing and facial flushing and periocular swelling observed in the 5-week study after the third dose coincident with the first appearance of ADAs. With the exception of emesis/vomitus, these clinical signs were effectively controlled with diphenhydramine pretreatment in the 5-week study and the subsequent 14-week study. There were no adverse SYNT001-related changes in weight gain, clinical chemistry, gross or histo-pathology. The No Observed Adverse Effect Level (NOAEL) was the highest dose tested in all 4 studies and the overall NOAEL following repeat weekly exposure to STYNT001 of up to 14 doses in cynomolgus monkeys was 100 mg/kg.

The safety, tolerability, and PD effect on total IgG levels in study SYNT-101—a Phase 1a study that assessed single ascending doses of SYNT001 in healthy male subjects—were also reviewed. In study SYNT-101, the doses of SYNT001 up to and including 30 mg/kg were well tolerated. There were no dose-limiting toxicities, serious adverse events (SAEs), or any other safety concerns. No adverse events (AEs) were observed in the 1 and 3 mg/kg dose cohorts. Headache was the most commonly reported treatment-emergent adverse event (TEAE), occurring in 8 of 11 subjects treated with 10 or 30 mg/kg SYNT001. One headache in the 10 mg/kg cohort was moderate (Grade 2) in severity; all other headaches were mild (Grade 1). One mild headache was treated with a single dose of acetaminophen; all other headaches resolved without treatment. Therefore, it is anticipated that the doses selected for this study should be well tolerated and have clinically relevant PD effects in patients with pemphigus.

Further consideration was given to the desired level of FcRn blockade to achieve suppression of IgG to a range that has been previously correlated with disease remission induced by immunoadsorption in autoimmune disorders such as pemphigus vulgaris and myasthenia gravis (ie, >50% decrease in total IgG from baseline) (Blaha et al., 2011; Eming and Hertl, 2006; Kohler et al., 2011).

The Sponsor also considered the potential effects of inhibiting FcRn function as they relate to IC associated innate and adaptive immunity. From the NHP studies, single doses of SYNT001 produced a dose-dependent decrease in total IgG and a further decrease was seen with repeated weekly doses up to a maximum 70% reduction at 100 mg/kg. This magnitude of total IgG reduction is approaching the expected maximal effect of 100% inhibition of FcRn function based on murine studies performed by the Sponsor and others (Nixon et al., 2015; Roopenian et al., 2003). In the recently completed Phase 1a trial with SYNT001 in healthy volunteers a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the NHP studies further reductions are expected following multiple dosing. A comparable

decrease in pathogenic autoantibodies is anticipated. In study SYNT-101, a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the NHP studies, further reductions may occur following multiple dosing.

For more information on the findings from the clinical and nonclinical findings with SYNT001, please refer to the Investigator's Brochure (IB).

### 2.3 Compliance Statement

This study will be conducted in compliance with Good Clinical Practice (GCP), including the International Conference on Harmonisation (ICH) Guidelines and FDA regulations, consistent with the principles outlined in the Declaration of Helsinki. In addition, the Investigator agrees to adhere to all applicable local laws and regulatory requirements relevant to the use of new therapeutic agents.

The study will be conducted in compliance with the protocol. The appropriate Institutional Review Boards (IRBs) must approve the protocol, any amendments, and the subject informed consent form (ICF) prior to implementation.

Freely given written informed consent must be obtained from every subject prior to participation in this clinical trial. As part of this procedure, the Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or AEs that may occur. The study subject should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The Investigator or designee will provide the Sponsor with a copy of the IRB-approved informed consent form prior to the start of the study. The rights, safety, and well-being of participating subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

#### 3. STUDY OBJECTIVES AND ENDPOINTS

#### 3.1 Primary Objective

The primary objectives of this study are as follows:

- Safety: To evaluate the safety of once-weekly IV infusions of SYNT001 at different dose levels and dosing durations in subjects with pemphigus (vulgaris or foliaceus)
- Dose Selection: To determine a Minimum Effective Dose (MED) of SYNT001 as assessed by (i) total IgG level nadir and (ii) the proportion of subjects that meet the criteria for response by Pemphigus Disease Area Index total activity score (PDAI)

#### 3.2 Secondary Objectives

The secondary objectives of this study are as follows:

- To determine the pharmacokinetics (PK) of SYNT001 following once-weekly IV infusions at different dose levels and dosing durations
- To evaluate the effect of once-weekly doses of SYNT001 at different dose levels and dosing durations on PD biomarkers
- To assess the effect of once-weekly doses of SYNT001 at different dose levels and dosing durations on disease markers
- To measure the immunogenicity of once-weekly doses of SYNT001 at different dose levels and dosing durations

#### 3.3 Exploratory Objectives

The exploratory objectives of this study are as follow:

- To explore the effect of once-weekly doses of SYNT001 at different dose levels and dosing durations on biomarkers to understand the pathophysiology of the disease and the SYNT001 mechanisms of action
- To determine the impact of different SYNT001 dose levels and dosing durations on the subject's use of corticosteroids to treat their pemphigus (vulgaris or foliaceus)
- To assess the impact of once-weekly doses of SYNT001 on the subject's health-related quality of life (HR-QoL) at different dose levels and dosing durations
- To assess the effect of once-weekly doses of SYNT001 on the appearance of skin and mucosal lesions at different dose levels and dosing durations
- To quantify the amount of SYNT001 in skin (skin biopsies optional)

#### 3.4 Primary Endpoints

The primary endpoints of this study are as follows:

Safety: The evaluation of SYNT001 safety based on vital signs, physical examinations, electrocardiograms (ECGs), clinical safety laboratory tests, the incidence of adverse events

(AEs), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) summarized by cohort, severity, and relationship to study product

Dose Selection: The determination of dose and dosing duration of SYNT001 that achieves (i) total IgG level nadir decrease by  $\geq$ 60% and  $\leq$ 90% from baseline and (ii) a PDAI total activity score of  $\geq$ 50% reduction from baseline to allow further clinical development in subject with pemphigus (vulgaris or foliaceus)

#### 3.5 Secondary Endpoints

The secondary endpoints of this study are as follows:

- The determination of PK parameters including half-life (t<sub>1/2</sub>), maximum serum concentration determined directly from the concentration-time profile (C<sub>max</sub>), observed time of peak plasma concentration (T<sub>max</sub>), area under the serum concentration-time curve from pre-dose (time₀) to 24 hours post-dose (AUC₀-2₄), and area under the serum concentration-time curve from pre-dose (time₀) to infinity (AUC₀-∞), (Cohort 1); maximum plasma concentration determined directly from the concentration-time profile (C<sub>max</sub>) and T<sub>max</sub> (Cohort 2 onwards) summarized by cohort and timepoint
- The evaluation of PD biomarkers based on absolute serum levels and percent change from baseline in serum levels of total immunoglobulin G (IgG), IgG subtypes (IgG1-4), immunoglobulin A (IgA), immunoglobulin M (IgM), albumin, and CIC summarized by cohort and timepoint
- The assessment of pemphigus disease activity by responses on PDAI based on absolute and percent change from baseline will be summarized by cohort and timepoint
- The assessment of pemphigus disease pathogenic antibody levels based on absolute and percent change from baseline of serum anti-desmoglein 1 and 3 antibody (anti-Dsg 1 and anti-Dsg 3) levels that will be summarized by cohort and timepoint
- The immunogenicity of once-weekly administered SYNT001 as determined by presence of anti-SYNT001 binding antibodies and neutralizing antibodies summarized by cohort and timepoint

### 3.6 Exploratory Endpoints

The exploratory endpoints of this study are as follows:

- The exploration of SYNT001 mechanisms of action and effects of SYNT001 on pathophysiology summarized by cohort and timepoint as determined by:
  - Complement component 3 (C3) levels by nephelometry
  - Anti-epithelial cell antibody (AECA) titers by indirect immunofluorescence
  - Fc gamma R2A receptor (FCGR2A) single-nucleotide polymorphisms (SNP) by genotyping
  - Presence of disease and inflammatory markers by RNAseq (RNA sequencing)
  - Immunophenotyping via measures of T cells, monocytes, NK cells and B cells by flow cytometry
  - Urine IgG levels to explore SYNT001 distribution and elimination

- Exploratory biomarkers to investigate immune response associated with pemphigus
- The evaluation of corticosteroid use during the study will be summarized by cohort and timepoint
- The assessment of SYNT001 impact on subject's HR-QoL by responses to the Autoimmune Bullous Disease Quality of Life (ABQoL) questionnaire and Skindex-29 scores summarized by cohort and timepoint
- The qualitative assessment of changes in appearance of skin and mucosal lesions as determined by photography presented by cohort and timepoint
- The determination of SYNT001 levels in skin biopsies across timepoints (skin biopsies optional)

Further details on the statistical and analytical plans for these endpoints are available in Section 11.

#### 4. STUDY DRUG

#### 4.1 Description of SYNT001

SYNT001 is provided in vials containing 5 mL SYNT001 (extractable volume) at a nominal concentration of 50 mg/mL. The product is supplied as a liquid at pH  $6.5 \pm 0.5$ . SYNT001 is diluted in dextrose 5% in water (D5W) to prepare the solution for infusion. SYNT001 will be infused via IV in 250 mL over 1 hour  $\pm$  15 minutes using a 0.2-micron, inline filter.

For detailed information regarding SYNT001 preparation and administration, refer to the Pharmacy Manual.

### 4.2 Dose Requirements

The specification for host cell deoxyribonucleic acid (DNA) in SYNT001 is <2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing per subject is limited to 5000 mg SYNT001.

For example, a subject with a body weight of 166 kg and enrolled in the ≤30 mg/kg dose cohort will receive ≤4960 mg SYNT001 per dose. If a subject's body weight extrapolates to an expected dose ≥5000 mg SYNT001, the dose will be capped to ensure the 5000 mg SYNT001 per dose limit is not exceeded.

A subject with a body weight of 111 kg and enrolled in the ≤45 mg/kg dose cohort will receive ≤4995 mg SYNT001 per dose. If a subject's body weight extrapolates to an expected dose ≥5000 mg SYNT001, the dose will be capped to ensure the 5000 mg SYNT001 per dose limit is not exceeded.

#### 4.3 Handling and Storage of SYNT001

All supplies of SYNT001 will be provided by the Sponsor and must be stored refrigerated (2°C to 8°C/36°F to 46°F) in the carton and protected from light, in a securely locked area, accessible to authorized persons only, until needed for dose preparation.

#### 4.4 Study Drug Accountability

The Investigator (or designee) is responsible for maintaining accurate accountability records of the study drug throughout the clinical study. Qualified site personnel will inventory the study drug received and will maintain records of disposition of the drug, including dates, quantity and use. All study drug received at the site must be accounted for on an accountability log provided by the Sponsor. All dispensing and accountability records will be available for Sponsor review. Study drug accountability will be verified during on-site monitoring visits.

Upon the completion or termination of the study, and upon written authorization from the Sponsor, or its representative, all unused and/or partially used study drug should be returned or destroyed at the investigational site, as specified by Sponsor. It is the Investigator's responsibility to ensure that the Sponsor, or its representative, has provided written authorization that procedures for proper disposal of the study drug have been established, and that appropriate

records of the disposal are documented and maintained. No unused study drug may be disposed of until fully accounted for by the Sponsor monitor (or designee).

#### 5. STUDY DESIGN

#### 5.1 Study Sites

This study will be conducted at approximately 10 global study sites.

#### 5.2 Overview of Study Design

This is a multicenter, open-label safety study to determine the dose regimen of SYNT001 administered intravenously in subjects with pemphigus (vulgaris or foliaceus). Approximately 20 (up to a maximum of 32) eligible subjects will receive planned doses of 10 mg/kg up to 45 mg/kg of SYNT001.

Cohorts will be dosed sequentially beginning with Cohort 1. Up to 8 eligible subjects will be enrolled in Cohort 1 and will receive 5 once-weekly 60-minute infusions of SYNT001 10 mg/kg. Based on review of safety, PD, and clinical outcomes of Cohort 1, sequential cohorts will enroll, pending recommendation received from a scheduled Dose Escalation Committee (DEC) review.

The DEC will consist of the Medical Monitor, an Independent Clinical Expert and a Syntimmune Medical Officer. To assist in the safety assessments, the DEC may request that Investigators, other experts, or members within their organization review the data and participate in the discussions.

Each cohort must be fully enrolled before a successive cohort will be opened for enrollment. An overview of the study cohorts is provided in Table 5 and Figure 1 shows a schematic of the study design.

**Table 5.** Cohort Overview

| Cohort No. | No. of Subjects | SYNT001 Dose | No. of Doses | DEC Review Timepoint |
|---|---|---|---|---|
| 1 <sup>a</sup> | up to 8 | 10 mg/kg | 5 | NA |
| 2 <sup>b</sup> | 4 <sup>c</sup> | ≤30 mg/kg <sup>d</sup> | 5 | When 100% of Cohort 1 subjects reach Day 42 |
| 3 <sup>b</sup> | 4° | ≤30 mg/kg <sup>d</sup> | 14 | When 50% of Cohort 2 subjects reach Day 42 |
| 4 <sup>b</sup> (optional) | 4 <sup>c</sup> | ≤45 mg/kg <sup>d</sup> | ≤14 | When 50% of Cohort 3 subjects reach Day 42 <sup>e</sup> |

Abbreviations: DEC = Dose Escalation Committee; NA = not applicable

- a. No more than 3 subjects with pemphigus foliaceus may be enrolled
- b. Two or fewer subjects with pemphigus foliaceus may be enrolled
- c. Up to 4 additional subjects may be added following DEC's evaluation.
- d. Dose will be recommended by the DEC and will be based on both an ongoing and set timepoint review of safety and pharmacodynamic evaluations including but not limited to, dose-limiting toxicities (DLTs), adverse events (AEs), treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and total IgG levels.
- e. All available data will be considered.

The first 2 subjects in Cohorts 1 and 2 will be enrolled at staggered intervals to facilitate adequate safety evaluation before dosing of subsequent subjects may proceed. A staggered

dosing interval for the first 2 subjects enrolled in successive cohorts will not be required if the planned dose is equal to or lower than that previously administered.

At 24-hour and 7-day intervals described below, the DEC will review of all available safety data (including but not limited to dose limiting toxicities [DLTs], AEs, TEAEs, and SAEs, PD (including but not limited to IgG levels), and clinical outcomes.

#### DEC Safety Review of 24-hour Data for Cohorts 1 and 2, Subject 1

The first 2 subjects will be dosed at least 24 hours apart. A DEC review of the 24-hour safety data for the first subject will be performed to ensure that there are no overt safety concerns before dosing the second subject.

#### Safety Review of 7-day Data for Cohorts 1 and 2, Subjects 1 and 2

The 7-day safety data for the first 2 subjects will be performed prior to dosing the remaining subjects in the cohort.

The 24-hour and 7-day reviews will consider seriousness and severity of AEs/TEAEs/SAEs and relatedness to study drug, vital sign assessments, physical examinations, and clinical laboratory testing.

For further information about dose escalation and study stopping rules, refer to Section 9.5.1 and Section 9.5.2, respectively.

#### 5.3 Randomization and Blinding

This is an open-label study.

#### 6. STUDY POPULATION

#### 6.1 Target Population

This study will be conducted in approximately 20 male and female subjects aged 18 and older with a confirmed diagnosis of pemphigus (vulgaris or foliaceus).

Up to 8 subjects may be enrolled in Cohort 1. Four subjects will be enrolled sequentially in Cohort 2, 3, and 4 (optional cohort). An additional 4 subjects may be enrolled in Cohorts 2, 3 and 4 (optional cohort) following DEC's evaluation and recommendation.

Subjects who withdraw for any reason other than an AE and who do not receive study drug or have only received one dose of study drug may be replaced, up to one subject per cohort. Thus, the maximum number of subjects who may be enrolled in this study is 36 (20 + up to 12 additional subjects, + up to 4 replacements, as necessary).

Within Cohort 1, no more than 3 subjects may be enrolled with pemphigus foliaceus. Within successive cohorts,  $\leq 2$  subjects with pemphigus foliaceus may be enrolled.

Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled visits.

#### 6.2 Inclusion Criteria

A subject must meet the following criteria to be eligible for the study:

- 1. Willing and able to read, understand, and sign an informed consent form.
- 2. Male or female  $\geq$ 18 years of age at the time of screening.
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/or skin lesions).
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal (ULN).
  - c. History of at least one positive tissue-based test (eg, biopsy, direct immunofluorescence [DIF]).
- 4. Active disease defined as lesions lasting >2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion >1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 mAb, last dose >12 months prior to screening.
  - b. If being treated with other immunosuppressants (ie, azathioprine, mycophenolate mofetil, methotrexate, dapsone, cyclosporine, tacrolimus, sirolimus, or low-dose cyclophosphamide [ $\leq$ 100 mg/day]), dose must be stable, defined as <25% change in dose, for 4 weeks prior to screening.
  - c. On stable dose of corticosteroids, defined as ≤1 mg/kg of prednisone or equivalent and may not be increased by more than 50% in the 2 weeks prior to screening.

- d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth.
- e. Stable use of topical low strength hydrocortisone ( $\leq 1\%$ ), tacrolimus, sirolimus, or pimecrolimus for lesions contributing < 10% of the PDAI total activity score for the 4 weeks prior to screening is allowed. Stable use of dexamethasone elixir solution (swish and spit only) for oral lesions for the 4 weeks prior to screening is allowed.
- f. If not on regular corticosteroids, no pulse corticosteroids are allowed in the 2 weeks prior to screening.
- 5. Body mass index (BMI)  $> 18.5 \text{ kg/m}^2$ .
- 6. Has a negative pregnancy test documented prior to the first dose of study drug (for women of childbearing potential).
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the screening period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 60 days after the final study visit.
- 10. A PDAI total activity score of >4 at screening.

#### 6.3 Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

- 1. Subject unable or unwilling to comply with the protocol.
- 2. Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ).
- 3. Positive for human immunodeficiency virus (HIV) or hepatitis C antibody.
- 4. Positive for hepatitis B surface antigen.
- 5. Active infection or history of recurrent infections.
- 6. IVIG treatment within 30 days of screening.
- 7. Received any cytotoxic (other than azathioprine) or any non-anti-CD20 mAb therapy in the 3 months prior to screening.
- 8. Any exposure to an investigational drug or device within the 30 days prior to screening.
- 9. Plasmapheresis or immunoadsorption within 30 days of screening.
- 10. Cellular therapy, including chimeric antigen receptor and T-cell (CAR-T), at any time prior to screening.
- 11. Use of any systemic or topical immunosuppressive drugs within 3 months of screening not including dose allowed by the inclusion criteria.
- 12. Serum total IgG <600 mg/dL.

- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (eg, a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results).
- 14. Any vaccination within 2 weeks of screening.

#### 7. STUDY PROCEDURES

#### 7.1 Informed Consent

All subjects must take part in the informed consent process. Adequate time must be allowed for the subject to ask questions and make a voluntary decision. No protocol-specific procedures, including screening procedures are to be performed until the subject has signed and dated an IRB-approved ICF. Subjects may withdraw consent at any time. Participation in the study may be terminated at any time without the subject's consent as determined by the Investigator.

### 7.2 Demographics and Medical History

Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and electronic case report form (eCRF). Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery, concomitant treatments, and relevant clinical response to past disease specific treatments including duration and dosing of such treatments.

### 7.3 Physical Examination

A complete physical examination will include measurements of weight (in kg) and height (in cm; height to be measured only at screening visit) and a review of the following body systems:

- General appearance
- Head, eyes, ears, nose, and throat
- Neck
- Respiratory
- Cardiovascular
- Abdomen
- Neurologic
- Extremities
- Dermatologic
- Lymphatic

Any abnormal and clinically significant findings from the physical examination must be recorded in the appropriate eCRF. Findings at screening and Day 0 (pre-dose) will be recorded as medical history.

### 7.4 Vital Sign Measurements

Vital sign assessments will include measurements of sitting blood pressure (mm Hg), heart rate (beats per minute), respiration rate (breaths per minute), pulse oximetry, and oral temperature (Celsius). Abnormal results are to be repeated after 5 minutes of rest. See Table 6 for timing window allowances with respect to measurement collection.

Vital sign measurements will be collected after the subject has been sitting for 5 minutes. Subjects should be seated quietly for at least 5 minutes in a chair with their backs supported, their feet flat on the floor (legs uncrossed), and their arms bared on a hard surface, with the arm slightly abducted and bent, with palm up and the midpoint of upper arm at heart level. Correct cuff and bladder size should be utilized and the same cuff and arm should be used per subject throughout study.

Vital sign measurements are to be obtained immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; 30 minutes, 1 hour, and 2 hours following completion of the infusion. Abnormalities in vital sign measurements will be graded in severity per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) scale Version 4.03.

Table 6. Timing Windows for PK/PD Sampling, ECG, and Vital Sign Measurements

| Time Point | Tolerance Window | |
|---|---|---|
| | Cohort 1 | Cohorts 2, 3, and 4<br>(Optional Cohort) |
| Pharmacokinetic Sampling | | |
| 0 hour | -240 minutes to 0 hour | -240 minutes to 0 hour |
| 5 minutes post end-of-infusion | ±5 minutes | ±5 minutes |
| 1 hour post end-of-infusion | N/A | ±15 minutes |
| 2 hours post end-of-infusion | ±15 minutes | ±15 minutes |
| 4 and 6 hours post end-of-infusion | ±15 minutes | N/A |
| 24 hours (1 day) post end-of-infusion | ±60 minutes | N/A |
| 48 hours (2 days) post end-of-infusion | $\pm 120$ minutes | N/A |
| Pharmacodynamic Sampling | | |
| 0 hour | -240 minutes to 0 hour | -240 minutes to 0 hour |
| 24 hours (1 day) post end-of-infusion | ±60 minutes | N/A |
| 48 hours (2 days) post end-of-infusion | $\pm 120$ minutes | N/A |
| ECG | | |
| 5 minutes post end-of-infusion | ±10 minutes | ±10 minutes |
| Vital Signs <sup>a</sup> | | |
| 0 hour | -240 minutes to 0 hour | -240 minutes to 0 hour |
| 15, 30, and 45 minutes after start of infusion | ±5 minutes | ±5 minutes |
| 1 hour after start of infusion | ±10 minutes | ±10 minutes |
| 30 minutes, 1 and 2 hours post end-of-infusion | ±10 minutes | ±10 minutes |

Abbreviations: ECG = electrocardiogram; N/A = not applicable; PD = pharmacodynamic; PK = pharmacokinetic.

a. Vital signs to include blood pressure, pulse rate, respiratory rate, oral temperature, and pulse oximetry.

### 7.5 Clinical Laboratory Measurements

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD samples, PK samples, and ADA samples) will be performed using established methods by a central laboratory. Clinical safety laboratory panels are listed in Table 7. Blood and urine samples for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and ADA samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Collection times for all safety, PD, and exploratory labs are outlined in Table 2, Table 3, and Table 4.

Table 7. Clinical Safety Laboratory Panels

| Hematology | Serum Chemistry | Urinalysis | Virology |
|---|---|---|---|
| <ul> <li>CBC with differential and blood smear</li> <li>Erythrocyte sedimentation rate</li> </ul> | <ul> <li>Albumin</li> <li>Alkaline phosphatase</li> <li>ALT</li> <li>AST</li> <li>BUN</li> <li>C-Reactive Protein</li> <li>Calcium</li> <li>Carbon dioxide</li> <li>Chloride</li> <li>Creatinine</li> <li>Glucose</li> <li>LDH</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total and direct bilirubin</li> <li>Total protein</li> <li>Uric acid</li> </ul> | <ul> <li>Appearance</li> <li>Color</li> <li>pH</li> <li>Specific gravity</li> <li>Ketones</li> <li>Protein</li> <li>Glucose</li> <li>Nitrite</li> <li>Urobilinogen</li> <li>Blood/hemoglobin</li> <li>Leukocyte esterase</li> <li>Bilirubin</li> <li>Microscopic examination of sediment: only if the results of the urinalysis dipstick evaluation are positive for blood/hemoglobin</li> </ul> | <ul> <li>Hepatitis C</li> <li>Hepatitis B</li> <li>HIV</li> <li>Tetanus</li> <li>VZV</li> </ul> |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; CBC = complete blood count; HIV = human immunodeficiency virus; LDH = lactate dehydrogenase; VZV = Varicella-Zoster virus.

Abnormalities in clinical laboratory tests that are considered clinically significant are to be recorded on the AE eCRF page. Laboratory results will be graded using the NCI CTCAE, Version 4.03. If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as an SAE (see Section 10.2.3).

For Cohort 1, the total blood draw for each subject who completes the study at Day 112 will be approximately 420 mL. For Cohort 2 the total blood draw for each subject who completes the study at Day 112 will be approximately 380 mL. For Cohort 3 and Cohort 4 (Optional), the total

blood draw for each subject who completes the study at Day 175 will be 656 mL. Please refer to the Laboratory Manual for more information.

#### 7.5.1 Pregnancy Testing

Pregnancy testing will be performed for women of childbearing potential. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.

#### 7.5.2 Virology

Testing for hepatitis C antibody, hepatitis B surface antigen, and HIV antibody will be performed at screening.

#### 7.5.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

Samples for serum tetanus antibody and VZV antibody testing are to be collected at baseline (pre-dose, Day 0), during the follow-up period, and at the end-of-study visit. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the protective level by the end-of-study visit, will be referred to their primary care physician for further management.

#### 7.5.4 Pharmacokinetics (PK) Sampling

The following PK parameters will be studied in Cohort 1:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-24}$ , and  $AUC_{0-\infty}$ . For all successive cohorts, the PK parameters studied will be  $C_{max}$  and  $T_{max}$ .

Specific collection times are detailed in Table 6. Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual

#### 7.5.5 Pharmacodynamic Sampling

PD samples will be collected for analyses throughout the study. Measurements for albumin will be derived from the clinical safety laboratory results. Specific collection times are detailed in. Samples for each type of PD will be collected according to the schedule shown in Table 8.
**Table 8.** Pharmacodynamic Assessments

| Parameter | <b>Collection Time Points</b> | | |
|---|---|---|---|
| | Cohort 1 | Cohort 2 | Cohort 3 |
| <ul><li>IgG</li><li>IgG subtypes (IgG1-4)</li><li>IgA</li><li>IgM</li></ul> | Screening and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, 56, 84, and 112 | Screening and Days 0, 7, 14, 21, 28, 35, 42, 56, 84, and 112 | Screening and Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 105, 119, 147, and 175 |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84, and 112 | Days 0, 7, 14, 21, 28, 35, 42, 56, 84, and 112 | Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 105, 119, 147, and 175 |
| Albumin | Screening and Days 0, 7, 14, 21, 28, 33, 42, 56, 84, and 112 | Screening and Days 0, 7, 14, 21, 28, 35, 42, 56, 84, and 112 | Screening and Days 0, 7,<br>14, 21, 28, 35, 42, 49, 56,<br>63, 70, 77, 84, 91, 98,<br>105, 119, 147, and 175 |
| Anti-Dsg (1 and 3) antibody titers | Screening and Days 0, 7, 14, 33, 56, 84, and 112 | Screening and Days 0, 7, 14, 21, 28, 35, 42, 56, 84, and 112 | Screening and Days 0, 7,<br>14, 21, 28, 35, 42, 49, 56,<br>63, 70, 77, 84, 91, 98,<br>105, 119, 147, and 175 |
| C3 and AECA levels<br>by indirect<br>immunofluorescence | Days 0, 14, 33, 56, 84, and 112 | Days 0, 35, and 56 | Days 0, 98, and 119 |
| Exploratory biomarkers (RNAseq, urine IgG) | Days 0, 14, 33, 56, 84, and 112 | Days 0, 35, and 56 | Days 0, 98, and 119 |
| Immunophenotyping<br>by flow cytometry for<br>measurement of T<br>cells, monocytes, NK<br>cells, and B cells | Days 0, 28, and 56 | Days 0, 35, and 56 | Days 0, 98, and 119 |
| Exploratory biomarker (FCGR2A SNP, via buccal swab) | Day 0 | Day 0 | Day 0 |
| Exploratory pemphigus immune response biomarkers | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84, and 112 | Days 0, 7, 14, 21, 28, 35, 42, 56, 84, and 112 | Days 0, 7, 14, 21, 28, 35, 42, 49, 56, 63, 70, 77, 84, 91, 98, 105, 119, 147, and 175 |

See Table 6 for timing window allowances with respect to measurement collection. More information, including detailed instructions for sample collection (including collection tubes) and preparation will be provided in a separate laboratory manual.

#### 7.5.6 Immunogenicity Testing

SYNT001 is being developed for the acute and chronic therapy of autoimmune disorders. Although SYNT001 is a humanized IgG4 mAb, exposure to SYNT001 in clinical trials could result in the development of ADAs, with potential consequences ranging from neutralization with possible lessening of drug efficacy to safety consequences such as allergic reactions. Testing will first detect binding ADAs. Then, for all confirmed positive samples, an ADA titer will be determined and there will be testing for neutralizing effects.

More information, including detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

# 7.6 12-Lead Electrocardiogram (ECG)

On dose administration days, digital 12-lead ECG measurements will be obtained at 5 minutes after the completion of the infusion. All ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each at an interval of 1 to 2 minutes apart. See Table 6 for timing window allowances with respect to performing ECG.

The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant.

Normal corrected QT interval using Fridericia's formula (QTcF) is ≤450 msec.

Abnormalities in the ECG that appear following therapy or that result in clinical signs and symptoms are considered clinically significant for the purposes of this study and will be recorded on the AE eCRF.

# 7.7 Pemphigus Disease Area Index (PDAI)

Pemphigus severity and disease activity will be measured using the PDAI in regions where a validated questionnaire is available. A PDAI total activity score will be determined at screening. To be eligible for study participation, the patient's grade by disease severity must be >4. Assuming subject eligibility, the PDAI will be administered during Treatment Period and Follow-up Period. Disease severity categories by PDAI are mild (0 to 8), moderate (9 to 24), and severe ( $\geq$ 25) (Shimizu et al., 2014). The Investigator will determine a PDAI score as follows: 0 to 250 points for disease activity ( $\leq$ 120 for skin,  $\leq$ 10 for scalp, and  $\leq$ 120 for mucosa), and 0 to 13 points for damage ( $\leq$ 12 for skin and  $\leq$ 1 for scalp) (Rosenbach et al., 2009). See Appendix 2.

### 7.8 Study Drug Administration

SYNT001 will be given as a 250-mL IV infusion over 1 hour  $\pm$  15 minutes using a 0.2-micron, inline filter.

#### 7.9 Photographs

Photographs will be taken of active lesions and follow-up photographs will be taken of the same areas at timepoints indicated in Table 2, Table 3, and Table 4. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

# 7.10 Health-Related Quality of Life Assessments

For Cohorts 2, 3 and 4 (optional cohort), health-related quality of life will be assessed using ABQoL and Skindex-29 in regions where a validated questionnaire is available. The ABQoL questionnaire was developed in Australia as a patient-based measure to quantify disease burden, monitor disease activity and evaluate response to therapeutic intervention in patients with autoimmune bullous disease (Sebaratnam et al., 2013; Sebaratnam et al., 2015) (Appendix 3). Skindex-29 was developed to measure the effects of skin disease on patients' quality of life using a self-administered 30 question dermatology survey (Chren et al., 1996) (Appendix 4).

#### 7.11 Adverse Event Assessments

Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form and continuing through the last study visit. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE. Clinical AEs will be graded using the NCI CTCAE, Version 4.03 (Appendix 1).

**Note:** AEs resulting in a subject's permanent discontinuation from the study, regardless of seriousness or relationship to study drug, MUST be promptly reported to the Sponsor. Additionally, subjects must be followed until return to normal and/or resolution of the AE.

See Section 10 for more information.

#### 7.12 Prior and Concomitant Medications

All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented on the source document and eCRF. A history of treatments taken for the primary disease, even if not taken within the 14 days prior to enrollment, will be collected.

#### **Permitted Medications**

Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not listed as prohibited.

- 1. Topical antibiotics to treat active infections that occur during the study.
- 2. Topical or systemic treatments for oral candidiasis.
- 3. Topical lidocaine for transient pain relief as needed.
- 4. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study.
- 5. Medication for potential infusion reactions: The Investigator may recommend prophylactic use of acetaminophen, IV hydration, diphenhydramine, histamine<sub>2</sub> (H<sub>2</sub>) blockers (eg, ranitidine, famotidine), etc to manage potential infusion reactions.
- 6. Low-strength corticosteroids (eg, hydrocortisone ≤1%) applied to a single lesion contributing <10% of the PDAI total activity score.
- 7. Topical tacrolimus, sirolimus or pimecrolimus applied to a single lesion contributing <10% of the PDAI total activity score.

 Syntimmune, Inc.

- 8. Dexamethasone elixir solution for oral lesions if dose remains stable throughout trial participation (swish and spit only).
- 9. Stable regimen of the following systemic immunosuppressants: azathioprine, mycophenolate mofetil, methotrexate, dapsone, cyclosporine, tacrolimus, sirolimus, or low dose oral cyclophosphamide (≤100 mg/day).

One month after the final dose of SYNT001, corticosteroids may be tapered at the Investigator's discretion.

#### **Prohibited Medications**

Use of the following medications will not be permitted during the study unless specified above as permitted:

- 1. Rituximab or other anti-CD20 antibody
- 2. Monoclonal antibodies other than study drug
- 3. Any topical or systemic immunosuppressive drugs apart from those that are listed as permitted.
- 4. IV corticosteroids prior to infusion (except in subjects who received corticosteroids for treatment of a prior infusion reaction to SYNT001)
- 5. Any dietary herbal supplements
- 6. Any investigational drug or device
- 7. Vaccinations within 2 weeks of screening through 28 days following final dose of study drug

# 7.13 Skin Biopsy

Optional skin biopsy samples from lesional or non-lesional skin will be collected to analyze SYNT001 levels.

#### 8. STUDY ASSESSMENTS

Study assessments are performed on a weekly basis and will be comprised of the following periods: Screening, Treatment (including Baseline [Day 0]), and Follow-Up (including End-Of Study). For those subjects that complete all periods in Cohorts 1 and 2, study duration is 112 days. For those subjects that complete all periods in Cohort 3, study duration is 175 days.

Further detail on specific study assessments is provided in Section 7.

# 8.1 All Cohorts: Screening Period and First Treatment (Day 0)

# 8.1.1 All Cohorts: Screening Period (Day -14 to Day -1)

For all cohorts, informed consent must be obtained before any study-specific samples are taken or study-specific tests or evaluations are conducted. The following assessments at the screening visit are to occur within 14 days before dosing. Study eligibility will be based on satisfying all the study inclusion and exclusion criteria (see Section 6).

At the screening visit, information will be collected and subjects will have clinical evaluations as follows:

- Informed consent
- Medical history and demographic data
- Review inclusion and exclusion criteria
- Complete physical examination, including height and weight
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- Hepatitis and HIV screen
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg1 and Dsg3 antibody titers
- Concomitant medication assessment
- AE assessment

#### 8.1.2 All Cohorts: Enrollment and First Treatment (Day 0)

For all cohorts, study Day 0 is defined as the date the subject is administered their first dose of study drug. On Day 0, subjects will be asked to come to the clinic and the following procedures will be performed prior to the first dose of study drug:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion

- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- Serum tetanus antibody and VZV antibody
- PDAI
- PK baseline sample collection (collected just prior to the start of the study drug infusion)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - FCGR2A SNP via buccal swab
  - RNAseq
  - Urine IgG
  - Immunophenotyping
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional) (Cohort 1 only)
- Photography
- HR-QoL assessments (ABQoL, Skindex-29) (Cohorts 2 and 3 only)

# After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest
- PK sample collection at 5 minutes. Thereafter at 2, 4, 6 hours (Cohort 1) or 1 and 2 hours (Cohorts 2 and 3) after the completion of study drug infusion; record collection date and time for each PK sample
- 12-lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion

#### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

## 8.2 Cohort 1: Day 1 to 84

# 8.2.1 Cohort 1: Follow-up Day 1

On Day 1 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Skin biopsy (optional)
- Concomitant medication assessment
- AE assessment

# 8.2.2 Cohort 1: Follow-up Day 2

On Day 2 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Skin biopsy (optional)
- Concomitant medication assessment
- AE assessment

#### 8.2.3 Cohort 1: Follow-up Day 5

On Day 5 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 0), subjects may return to the clinic or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment

## 8.2.4 Cohort 1: Treatment Day 7 (Dose 2)

On Day 7 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - Exploratory pemphigus immune response biomarkers

# After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

#### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

#### 8.2.5 Cohort 1: Follow-up Day 12

On Day 12 ( $\pm$  6 hours), subjects may return to the clinic or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers

- If visit performed at the study site: 12-lead ECG to be obtained in triplicate
- Concomitant medication assessment
- AE assessment

# 8.2.6 Cohort 1: Treatment Day 14 (Dose 3)

On Day 14 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

#### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

## 8.2.7 Cohort 1: Follow-up Day 19

On Day 19 ( $\pm$  6 hours), subjects may return to the clinic or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment.

# 8.2.8 Cohort 1: Treatment Day 21 (Dose 4)

On Day 21 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

#### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### 8.2.9 Cohort 1: Treatment Day 28 (Dose 5)

On Day 28 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PK sample collection (collected just prior to the start of the study drug infusion)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Immunophenotyping
  - Exploratory pemphigus immune response biomarkers

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest
- PK sample collection at 5 minutes and 2, 4, and 6 hours after the completion of study drug infusion; record collection date and time for each PK sample
- 12-lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion

#### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

#### **8.2.10** Cohort 1: Follow-up Day 29

On Day 29 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment
- AE assessment

# **8.2.11** Cohort 1: Follow-up Day **30**

On Day 30 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment
- AE assessment

# 8.2.12 Cohort 1: Follow-up Day 33

On Day 33 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 28), subjects will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers

 Syntimmune, Inc.

- Skin biopsy (optional)
- Photography
- Concomitant medication assessment
- AE assessment

# 8.2.13 Cohort 1: Follow-up Day 42

On Day 42 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment

# 8.2.14 Cohort 1: Follow-up Day 56

On Day 56 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position)
- Serum tetanus antibody and VZV antibody
- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Immunophenotyping

- Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)
- Photography
- Concomitant medication assessment
- AE assessment.

### 8.2.15 Cohort 1: Follow-up Day 84

On Day 84 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Serum tetanus antibody and VZV antibody
- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)
- Photography
- Concomitant medication assessment
- AE assessment

Note: Cohort 1 End-of-Study visit is detailed in Section 8.4.

# 8.3 Cohorts 2 and 3: Subsequent Treatments to Follow-up

# 8.3.1 Cohort 2: Treatment Days 7 and 21; Cohort 3: Treatment Days 7, 14, 21, 28, 35, 49, 56, 63, 70, 77, and 84

For Cohort 2 Days 7 and 21 ( $\pm$  1 day) and Cohort 3 Days 7, 14, 21, 28, 35, 49, 56, 63, 70, 77, and 84 ( $\pm$  1 day), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

 Syntimmune, Inc.

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - Exploratory pemphigus immune response biomarkers

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

## Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

# 8.3.2 Cohort 2: Treatment Days 14 and 28; Cohort 3: Treatment Days 42 and 91

For Cohort 2 Days 14 and 28 ( $\pm$  1 day) and Cohort 3 Days 42 and 91 ( $\pm$  1 day), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test (Cohort 3, Days 42 and 91 only)
- PDAI
- PK sample collection (collected just prior to the start of the study drug infusion) (Cohort 2, Day 28 only; Cohort 3, Day 91 only)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)

- IgG, IgG subtypes (IgG1-4), IgA, IgM
- CIC
- Anti-Dsg (1 and 3) antibody titers
- Exploratory pemphigus immune response biomarkers
- Photography (Cohort 3, Day 42 only)

#### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest
- PK sample collection at 5 minutes and 1 and 2 hours after the completion of study drug infusion; record collection date and time for each PK sample (Cohort 2, Day 28 only; Cohort 3, Day 91 only)
- 12-lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion

#### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### 8.3.3 Cohort 2: Follow-up Days 35 and 56; Cohort 3: Follow-up Days 98 and 119

For Cohort 2 Days 35 ( $\pm$  1 day) and 56 ( $\pm$  3 days) and Cohort 3 Days 98 ( $\pm$  1 day) and 119 ( $\pm$  3 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test (Cohort 2, Day 56 only; Cohort 3, Day 119 only)
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Cohort 2, Day 56 only; Cohort 3, Day 119 only)
- Serum tetanus antibody and VZV antibody (Cohort 2, Day 56 only; Cohort 3, Day 119 only)
- PDAI
- Immunogenicity sample collection (Cohort 2, Day 56 only; Cohort 3, Day 119 only)
- PD sample collection

- IgG, IgG subtypes (IgG1-4), IgA, IgM
- CIC
- Anti-Dsg (1 and 3) antibody titers
- C3
- AECA
- RNAseq
- Urine IgG
- Immunophenotyping
- Exploratory pemphigus immune response biomarkers
- Photography
- HR-Qol (ABQoL, Skindex-29)
- Concomitant medication assessment
- AE assessment

## 8.3.4 Cohort 2: Follow-up Days 42 and 84; Cohort 3: Follow-up Days 105 and 147

For Cohort 2 Days 42 ( $\pm$  1 day) and 84 ( $\pm$  5 days) and Cohort 3 Days 105 ( $\pm$  1 day) and 147 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - \_ CIC
  - Anti-Dsg (1 and 3) antibody titers
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment

# 8.4 All Cohorts: End of Study or Early Termination Visit; Cohorts 1 and 2, Day 112; Cohort 3, Day 175

For Cohorts 1 and 2 Day 112 ( $\pm$  5 days) and Cohort 3 Day 175 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- Serum tetanus antibody and VZV antibody

- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3 (Cohort 1 only)
  - AECA (Cohort 1 only)
  - RNAseq (Cohort 1 only)
  - Urine IgG (Cohort 1 only)
  - Exploratory pemphigus immune response biomarkers
- Photography
- HR-Qol (ABQoL, Skindex-29) (Cohorts 2 and 3 only)
- Concomitant medication assessment
- AE assessment

**Note**: a subject may choose to terminate participation in the study at any time. Under this circumstance, the subject will be encouraged to return as soon as possible for an early treatment visit and to receive assessments otherwise scheduled on Day 112 (Cohorts 1 and 2) or Day 175 (Cohort 3).

# 9. STUDY RULES

# 9.1 Subject Withdrawal

Every reasonable effort will be made to keep the subject in the study; however, if a subject withdraws from the study, the Investigator should complete and report the reasons for withdrawal as thoroughly as possible. The reason(s) for termination must be clearly documented on the appropriate page of the eCRF.

If a subject discontinues from the study for any reason, every effort will be made to collect all clinical and laboratory data as scheduled for the Early Termination Visit (see Section 8.4). If the subject fails to return for these assessments for unknown reasons, every effort (eg, telephone, email, and letter) should be made to contact them.

The reason(s) for a subject's participation in the study may be prematurely discontinued will be documented and include:

- 1. The subject wishes to withdraw from the study.
- 2. Request by a regulatory agency (eg, Institutional Review Board).
- 3. The subject experiences a significant or intolerable AE.
- 4. The subject experiences a significant adverse change in vital signs, physical examination findings, or clinical laboratory parameter.
- 5. The subject has a need for a concomitant medication that is not permitted by the study protocol.
- 6. The subject experiences generalized impairment or mental incompetence that would result in the subject being unable to understand his or her participation in the study.
- 7. If, in the Investigator's medical judgment, further participation would be injurious to the health and well-being of the subject, or is not in the best interest of the subject.
- 8. Administrative reasons, such as subject non-compliance or a major protocol violation.
- 9. The subject requires a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus (at the discretion of the Investigator with consultation with the Medical Monitor).

If at the discretion of the Investigator with consultation with the Medical Monitor, a subject requires a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus, the subject will be encouraged to continue their study visits to allow collection of safety data.

### 9.2 Subject Replacement

Enrolled subjects withdrawn for a reason other than an AE will be replaced if they have not been dosed or have only received one dose of study drug at the time of discontinuation, up to one subject per cohort. Subjects who do not receive all doses of study drug will continue to be followed through all scheduled study visits.

# 9.3 Study Discontinuation

The Sponsor has the right to terminate or to stop the study at any time. Reasons for study discontinuation may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other related studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Drug supply issues
- Excessive subject self-withdrawal
- Significant protocol violations (eg, violation of eligibility criteria, dosing errors, missing data for study endpoint analysis)

# 9.4 Lost to Follow-up

All reasonable effort should be made to contact any subject lost to follow-up during the study to complete assessments and retrieve any outstanding data. If the subject is unreachable after three good faith attempts, at a minimum, the Investigator should follow up with a registered letter requesting contact so safety data may be collected, recorded, and reported (if necessary).

#### 9.5 Stopping Rules

# 9.5.1 Dose-Escalation Stopping Rule

Dose recommendations will be made by a DEC based upon a review of all available safety data, on a continuous basis as well as at discrete timepoints. Available data will be based on safety and pharmacodynamic evaluations including but not limited to, DLTs, AEs, TEAEs, SAEs, PD (including but not limited to IgG levels), and clinical outcomes.

Dose-limiting toxicity (DLT) will be defined generally as severe (Grade 3) AEs occurring in ≥2 subjects in any cohort that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. Upon review of the available information, the DEC may reduce the dose prior to enrolling additional subjects using the guidelines below:

- Cohort 1: Dose may be reduced by at least 50%.
- Cohort 2: Dose may be reduced by at least 33%.
- Cohort 3: Dose may be reduced to a level lower than the Cohort 2 dose.
- Cohort 4 (optional cohort): Dose may be reduced to level lower than the Cohort 3 dose.

# 9.5.2 Study Stopping Rule

If any subject experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, any further dosing in all enrolled subjects will be suspended until the DEC has evaluated the event and determined the next appropriate course of action. At any time during the study, the study may be discontinued if the DEC determines that further drug exposure would pose an undue risk to subjects.

# 9.5.3 Individual Stopping Rule

Dosing for any individual subject will be discontinued (ie, no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related non-serious AE that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) suggest that it could be unsafe to administer further study drug to that subject.

Subjects who are withdrawn from this study due to an AE determined to be related to study drug are to be followed until there is:

- Resolution or stabilization of the AE determined to be related
- The subject is lost to follow-up
- The event is otherwise explained

If there is a persistent AE contributing to discontinuation that is determined to be related to SYNT001, subjects must be followed with appropriate medical management until resolution or stabilization. Refer to Section 10 for more information.

### 10. EVALUATION OF SAFETY

# **10.1** Safety Parameters

Subjects will be monitored continuously throughout the treatment and follow-up period for AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status. Parameters measure/assess safety include physical examinations, vital sign measurements (including pulse oximetry), clinical (safety) laboratory tests (hematology, serum chemistries, urinalysis), concomitant medication assessments, and ECG. Clinical and laboratory AEs will be graded using the NCI CTCAE; Version 4.03 (see Appendix 1).

#### 10.2 Adverse Events

An AE is defined as any untoward medical occurrence in a clinical trial subject associated with the use of a drug, whether considered drug related or not. An AE can be an unfavorable and unintended sign (eg, an abnormal laboratory value finding), a symptom, or a disease temporally associated with the use of a drug, without judgment as to causality. An AE can arise from use of the drug (eg, use in combination with another drug) and from any route of administration, formulation or dose, including an overdose. An AE also includes, but is not limited to, any clinically significant worsening of a pre-existing condition. Examples include:

- Any sign, symptom, physical finding, or laboratory result that has worsened in nature, severity or frequency compared to baseline
- Reactions from an investigational drug, including those occurring because of an overdose, abuse of the study drug, withdrawal phenomena, sensitivity or toxicity
- Concurrent illness that was not present or worsens in nature, severity, or frequency compared to baseline
- Injury or accident
- Exacerbation of a pre-existing condition

Pregnancy is not considered an AE or SAE; however, any pregnancy complication(s) should be recorded as an AE(s) or SAE(s) (if applicable). Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions. Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. If a female subject becomes pregnant during the conduct of the study, the Investigator must notify the Sponsor according to the procedures provided in Section 10.5.4.

Planned hospitalization admissions or surgical procedures for a condition known to exist before the subject signed the informed consent are not an AE and should be recorded as medical history. If the planned hospitalization or procedure is executed as planned and without complication, the record in the subject's medical history is considered complete. However, if the event/condition deteriorates in an unexpected manner during the study or following surgery, it must be reported as an AE according to the procedures provided in Section 10.2.1.

#### 10.2.1 **Recording an Adverse Event**

For data collection, all untoward events that occur after informed consent through the last study visit are to be recorded on eCRFs by the investigational site. All AEs are to be accurately recorded on the Adverse Event page of the subject's eCRF. The severity of each AE will be graded using the NCI CTCAE, Version 4.03 (see Appendix 1). The date of onset as well as the end date of the event should be recorded or the event should be entered as "ongoing". In addition, the method used to treat the AE and the outcome of the AE will be noted. The Investigator will assess the relationship of the event to study drug.

#### 10.2.2 **Assessment of Causality**

A medically qualified Investigator must assess the relationship of any AE (including SAEs) to the use of the study drug, as related or not related, based on clinical judgment and using all available information. The causal relationship between the study medication and the AE will be assessed using one of the following categories:

**Not Related:** Factors consistent with an assessment of Not Related include:

- Temporal relationship is lacking (eg, the event did not occur within a reasonable time frame following administration of the study medication); or
- Other causative factors more likely explain the event (eg, a pre-existing condition, other concomitant treatments).

**Related:** Factors consistent with an assessment of Related include:

- There is a positive temporal relationship (eg, the event occurred within a reasonable time frame following administration of study medication); or
- The AE is more likely explained by the investigational product than by another cause (ie, the AE shows a pattern consistent with previous knowledge of the investigational product or the class of the investigational product)

#### 10.2.3 **Serious Adverse Events**

(Notify Medpace Safety within 24 hours; document on eCRF)

The SAE definition and reporting requirements are in accordance with Title 21 Part Code of Federal Regulations (CFR) 312.32 and the Guidance for Industry and Investigators Safety Reporting Requirements for Investigational New Drug (INDs) and Bioavailability /Bioequivalence Studies.

An AE is considered "serious" if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:

**Death:** This includes any death that occurs while the subject is "on study" through the last study visit.

 Syntimmune, Inc.

- <u>Life-threatening adverse drug event:</u> An AE or suspected adverse reaction is considered "life threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.
- <u>Inpatient hospitalization or prolongation of existing hospitalization:</u> an AE that requires admission to a hospital for medical and/or surgical intervention.
  - In the absence of an AE, the Investigator should <u>not</u> report hospitalization or prolongation of hospitalization as an SAE, as detailed in the following examples:
    - An elective or previously scheduled surgery for a pre-existing condition that has not deteriorated unexpectedly after initiation of treatment (eg, a previously scheduled ventral hernia repair)
    - Hospitalization or prolongation of hospitalization is needed for a procedure required by the protocol
    - Hospitalization or prolongation of hospitalization is part of routine procedure followed by study center
    - o Hospitalization for survey visits, annual physicals, or planned observation
    - Hospitalization for observation with release within 24 hours (eg, an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Congenital anomaly/birth defect
- <u>Important medical event:</u> An event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### **10.2.3.1** Recording a Serious Adverse Event

When the diagnosis of an SAE is known or suspected, the Investigator should record the diagnosis or syndrome as the primary SAE term, rather than as signs or symptoms. Signs and symptoms may then be described in the event description. For example, dyspnea should not be used as an SAE term if the diagnosis, which caused the dyspnea, is known to be malignant pleural effusion.

Death should not be recorded as an SAE, but as an outcome of a specific SAE, unless the event preceding the death is unknown. In the exceptional case where the events leading to death are unknown, then death may be used as an event term. If an autopsy was performed, the autopsy the autopsy report should be provided.

#### 10.2.3.2 Reporting a Serious Adverse Event

#### RESPONSIBILITIES OF THE INVESTIGATOR

Any death, SAE, or pregnancy, experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the Sponsor (or designee).

Contact information for SAE reporting:



Additionally, the Investigator will be able to contact the **Medical Monitor**:

# **Medical Safety Contact**



The Investigator will report the SAE to his or her IRB in accordance with IRB's standard operating procedures and policies. Adequate documentation must be maintained showing that the IRB was properly notified.

SAEs must be recorded on the SAE form in the electronic data capture (EDC) system. This requirement includes all SAEs that occur after informed consent through the last study visit. The minimum information required for SAE reporting includes identity of investigator, site number, subject number, an event description, SAE term(s), onset date, the reason why the event is serious (ie, the seriousness criteria), and the Investigator's assessment of the relationship of the event to study treatment. Additional SAE information including medications or other therapeutic measures used to treat the event, action taken with the study treatment due to the event, and the outcome/resolution of the event will be recorded. Paper forms for reporting SAEs will be provided to the study sites as back-up in case the EDC system is not accessible.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. Furthermore, the Investigator may be required to provide supplementary information as requested by the Sponsor (or designee).

#### RESPONSIBILITIES OF THE SPONSOR (OR DESIGNEE)

The Sponsor (or designee) will process and evaluate all SAE as soon as the reports are received. For each SAE received, the Sponsor will decide as to whether the criteria for expedited reporting have been met.

The Sponsor (or designee) is responsible for promptly informing the FDA and other regulatory authorities as well as other participating Investigators of the event. Written submission must be made by the Sponsor to the FDA as soon as possible and in no event later than 15 calendar days after the Sponsor's initial notification of the event, or for an event that is fatal or life-threatening no later than 7 calendar days after the Sponsor's initial notification.

#### **EXPEDITED REPORTING**

Under FDA ruling (US Code of Federal Regulations, Title 21 CFR Part 312.32) and the ICH Guideline "Clinical Safety Data Management: Definitions and Standards for Expedited Reporting E2A," the Sponsor is required to submit written documentation, in the form of a safety report, detailing:

- Any event associated with the use of the drug, that is both serious and unexpected, or
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects, including reports of mutagenicity, teratogenicity, or carcinogenicity.

The Sponsor will submit SAEs that meet the criteria for expedited reporting to the regulatory authorities in accordance with local regulations governing safety reporting.

#### 10.2.4 Follow-Up of Adverse Events and Serious Adverse Events

Any SAE or AE must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. Appropriate diagnostic tests should be performed and therapeutic measures, if indicated, should be instituted until the event has returned to baseline or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary. The status of all AEs will be documented as of the last study visit. If all required information is not available at the time of the initial report, follow-up information will be completed in the EDC system.

# 10.3 Warnings and Precautions

#### 10.3.1 Vaccinations

Subjects must not receive any vaccinations from within 2 weeks of screening until 28 days following final dose at the discretion of the Investigator.

## 10.3.2 Management of Allergic or Infusion-Related Reactions

As observed with all mAbs administered by IV infusion, infusion reactions to SYNT001 are possible. In general, infusion reactions to mAbs observed in human studies typically develop

 Syntimmune, Inc.

within 30 minutes to 2 hours after the initiation of drug infusion, although symptoms may be delayed for up to 24 hours. These infusion reactions can occur with the first dose of a mAb and are generally mild in severity, although severe and even fatal reactions can occur.

Allergic and/or infusion-related reactions include hypersensitivity reactions and cytokine release syndromes. These reactions are experienced by subjects during or within hours of the infusion of mAb therapy. Symptoms can include flushing, alterations in heart rate and blood pressure, dyspnea, bronchospasm, back pain, fever, urticaria, edema, nausea, and all types of rashes. Anaphylaxis is recognized as a severe, life-threatening, generalized, or systemic reaction. This is a medical emergency characterized by rapidly developing life-threatening airway and/or breathing and/or circulation problems usually associated with skin or mucosal changes.

Management of Grade 1 infusion reactions include interrupting the infusion or decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone, or acetaminophen, either alone or in combination, depending on the subject's signs and symptoms. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 preparation.

Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. Continued treatment with SYNT001 is prohibited following Grade 2 or higher infusion reactions. See Figure 2 and Figure 3 for details on the management of Grade 2 and Grade 3 infusion reactions. Allergic or infusion-related reactions will be graded in severity and managed based on NCI CTCAE Version 4.03 (see Table 9).

Figure 2. Management of Moderate (Grade 2) Infusion Reactions



If symptoms and signs resolve completely either spontaneously or after administration of diphenhydramine with or without hydrocortisone, consider rechallenge:

Wait at least 20 minutes following medication administration before commencing rechallenge at an infusion rate of 50% or less of the initial infusion rate or

Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 administration.

Figure 3. Management of Severe (Grade 3 or Higher) Infusion Reactions

Subject presents with any of the below:

- Urticaria
- Airway threatened by angioedema
- Angioedema: Lip, mouth, facial swelling
- Respiratory compromise wheezing, dyspnea, stridor or hypoxia (O<sub>2</sub> saturation <90%)</li>
- BP <90 mmHg SBP or >30% decrease from patient baseline



Start basic life support:

- High oxygen flow
- On bed, head down, legs up
- Large bore IV cannula, 1 L normal saline STAT
- Initiate vital signs at least every 15 minutes



Consider (under medial direction):

Epinephrine 1:1000

• 0.3 mg (0.3 mL) IM into lateral thigh



Airway Threatened: Nebulized epinephrine 1:1000, 3–5 mL (3–5 mg)

**Bronchospasm:** Nebulized salbutamol 5 mg

(Wheeze or Hypoxia) Consider: Intubation / nebulized epinephrine

**Hypotension:** Place on cardiac monitor

(Systolic BP <100 mmHg) Further epinephrine 1:1000, 0.3 mg IM and

IV normal saline bolus 20 mL/kg STAT as needed

Have vasopressin on hand



Transfer to Emergency Room/ICU Observe until all symptoms resolved.

Table 9. Grading and Management of Allergic or Infusion-Related Reactions

| Adverse | Grade | | | | |
|---|---|---|---|---|---|
| Event | 1 | 2 | 3 | 4 | 5 |
| Infusion-<br>related<br>reaction | Mild transient<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤24 hours | Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Allergic reaction | Transient<br>flushing or<br>rash, drug<br>fever<br><38.0°C.<br>Intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤24 hours | Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (eg, renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Anaphylaxis | _ | _ | Symptomatic<br>bronchospasm, with or<br>without urticarial;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Cytokine<br>release<br>syndrome | Mild reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤24 hours | Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (eg, renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>pressor or<br>ventilator<br>support<br>indicated | Death |

Abstracted from NCI CTCAE Version 4.03.

#### **10.3.3** Potential Immune Effects

An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels after a single dose and further decreases after multiple doses up to a 70% to 80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will

occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within 30% of baseline levels observed at pretreatment occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.

Given the normal adult range of total IgG of 500 to 1600 mg/dL (Agarwal and Cunningham-Rundles, 2007; Furst, 2009; Gonzalez-Quintela et al., 2008; Jolliff et al., 1982; Keystone et al., 2007; McMillan et al., 1997; van Vollenhoven et al., 2013), with a mean of 1150 mg/dL, a 50% decrease in the mean would be to 575 mg/dL and a 50% decrease from the low end of the normal range used for the inclusion criteria of 600 mg/dL in this study would be to 300 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 120 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency (Ameratunga et al., 2013), the levels will be transient. Further, as reported for other therapies used for pemphigus, the temporary (ie, less than 4 months) depletion of IgG (up to 95% reduction of total IgG as seen with immunoadsorption) does not appear to impart an increased risk of infection (Eming and Hertl, 2006; Furst, 2009; Keystone et al., 2007; Schmaldienst et al., 2001; van Vollenhoven et al., 2013). Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to reverse the low IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

An antibody that blocks FcRn is expected to also down-modulate innate and adaptive immunity and the catabolism of IgG-containing immune complexes (IC). Specifically, it is expected that anti-FcRn will promote the clearance of IgG-containing ICs and the effects of these ICs on stimulating innate immune cell production of inflammatory cytokines (eg, interleukin 12 [IL-12], interferon-γ, and tumor necrosis factor [TNF]) and inhibit the processing and presentation of antigens contained within ICs and thus the antigen-specific activation of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells. Therefore, subjects with pre-existing conditions that are dependent upon IgG antibodies, such as chronic infections (eg, HIV, HBV or HCV), will be excluded from this study, as will subjects with active infection, in general.

### **10.4** Events of Special Interest

Not applicable.

#### 10.5 Other Safety Considerations

#### 10.5.1 Laboratory Data

All laboratory data obtained during the study should be reviewed. Any abnormal value that leads to a change in subject management (eg, requirement for additional medication or monitoring) or is determined to be of clinical significance by the Investigator should be reported as an AE and/or SAE as appropriate, unless this value is consistent with values obtained before entry into the study.

#### 10.5.2 **Medication Errors**

Any medication error that results in an AE, even if it does not meet the definition of serious, requires reporting within 24 hours to the safety Medical Monitor. Refer to Section 10.2.3.2 for more information.

#### 10.5.3 Overdose

For the purposes of this study, an overdose of SYNT001 is defined as a dose that is two-fold higher than the intended dose for the subject. As all dosing for this study will be conducted in a controlled clinical setting, an overdose is not anticipated. In the unlikely event an overdose should occur, it should be reported as an AE.

#### 10.5.4 **Pregnancy**

If a female subject or the female partner of a male subject becomes pregnant during the course of the study, the Investigator must report the pregnancy to Medpace Safety using the **Pregnancy Reporting Form** within **24 hours** of becoming aware of the event. The Investigator must obtain consent to collect pregnancy information (including the status of the newborn, if applicable).

If some of the information required for completion of the Pregnancy Reporting Form is unavailable at the time of the initial report, follow-up reports will be completed and submitted within 24 hours of becoming aware of the new information. Any pregnancy will be followed through delivery for the observation of any SAEs. Any SAE that occurs during pregnancy must be recorded on the SAE report form in the EDC system (eg, maternal serious complications, therapeutic or spontaneous abortion, ectopic pregnancy, stillbirth, neonatal death, congenital abnormality, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs (see Section 10.2.3.2).

### 11. STATISTICAL CONSIDERATIONS

# 11.1 General Design

This study is being conducted to evaluate the safety, tolerability, PK, PD, activity, and immunogenicity of SYNT001 in pemphigus patients.

#### 11.2 Study Populations

Three populations will be employed in the analysis of study data:

- The **Safety** population will consist of all subjects who have received at least one dose of study drug.
- The **PD** population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.
- The **PK** population will consist of all subjects who receive at least one dose of study drug and have post-dose PK data available.

Primary safety analyses will be performed on the safety population. Demographics, subject disposition, screening, and baseline characteristics will be summarized for the safety and PD/PK populations, where appropriate.

# 11.3 Sample Size Justification

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

### 11.4 Statistical Analysis

#### 11.4.1 Statistical Analysis Plan

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). The SAP may modify the plans outlined in the protocol; however, any deviations from the previously approved statistical plan will be described and justified in a SAP amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate and will be described in the SAP. The SAP including pharmacokinetic data analysis methodologies will be finalized prior to database lock.

All descriptive and inferential statistical analyses will be performed using Statistical Analysis System (SAS) version 9.4 or later. Missing data will not be imputed unless otherwise stated. All clinical data captured will be provided in data listings.

Methods of handling of missing data for different endpoints will be further specified in the SAP. In general, where individual data points are missing because of insufficient samples, dropouts, or other reasons, the data will be analyzed based on reduced denominators unless specified otherwise in the SAP.

#### 11.4.2 Statistical Methodology

All clinical data captured will be provided in data listings. Subject disposition, demographic information, and baseline characteristics will be presented. Baseline will be defined at the last value obtained prior to the first dose of study drug. Results will be summarized by dose level and cohort. Any discrepancy between treatment to be given and treatment received will be accounted for in these displays.

Continuous data will be summarized using descriptive statistics: number of subjects (N), number of observations (n), mean, median, standard deviation (SD), minimum, and maximum.

Categorical data will be summarized using frequencies and percentages. When categorical data will be presented, the percent will be suppressed when the count is zero to draw attention to the non-zero counts. The denominator for all percentages, unless otherwise specified, will be the number of subjects in the specified analysis population.

# 11.4.3 Analysis of Primary Endpoints

#### **11.4.3.1** Safety Data

All statistical analysis of safety outcomes will be descriptive. Safety observations and measurements include AEs, treatment-emergent AEs (TEAEs), SAEs, clinical safety laboratory tests, vital sign measurements, physical examinations, and ECGs. The incidence of AEs, TEAEs and SAEs will be summarized by cohort, severity and relationship to study product.

TEAEs will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least one occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study treatment) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject, dose, and overall per SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by cohort and time point. The incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the local laboratory.

Vital sign measurements and change from baseline will be summarized at each scheduled time point by cohort using descriptive statistics.

Arithmetic mean of parameters from triplicate ECG will be calculated first for each subject at each planned time point. Then summary statistics of ECG test parameters (mean of triplicate) and change from baseline to each post-dose time point will be calculated. Shift tables for ECG test result category change (normal, abnormal, clinically abnormal) from pre-dose to each post-dose time point showing number and percentage of subjects with movement between categories

will be presented by treatment group. Frequency and percentage of subjects experiencing potential QTc prolongation (QTcF > 450) will be summarized at each time point by cohort.

Concomitant medications will be coded using WHO Drug Dictionary (WHO-DD March 2013, Type B2 or later) and the data will be summarized and presented in tables and listings.

#### 11.4.3.2 Dose Selection Data

The evaluation of SYNT001 based on total IgG levels and responses on the PDAI total activity score from baseline will be summarized using descriptive statistics. Descriptive statistics will include mean, SD, coefficient of variation (CV), median, minimum, and maximum. The determination of dose and dosing duration of SYNT001 that achieves (i) total IgG level nadir decrease by  $\geq$ 60% and  $\leq$ 90% from baseline and (ii) a PDAI total activity score of  $\geq$ 50% reduction from baseline to allow further clinical development in subject with pemphigus (vulgaris or foliaceus).

# 11.4.4 Analysis of Secondary Endpoints

#### 11.4.4.1 Pharmacokinetic Data

PK results for SYNT001 will be summarized by cohort and timepoint.

Study drug serum concentrations will be used to calculate the following PK parameters: t<sub>1/2</sub>, C<sub>max</sub>, T<sub>max</sub>, and AUC<sub>0-24</sub> and AUC<sub>0-∞</sub> in Cohort 1 and C<sub>max</sub> for Cohorts 2, 3, and 4 (optional cohort). PK parameters will be determined using noncompartmental method(s). Descriptive statistics will be provided for the PK parameters including mean, SD, CV, median, minimum, and maximum. T<sub>max</sub> will be reported as median and range. All descriptive statistics will be performed on untransformed PK parameters and after log<sub>10</sub> transformation of PK parameters.

For calculation of mean concentrations and generation of mean concentration-time profiles, all below the limit of quantification (BLQ) values will be set to zero except when an individual BLQ falls between 2 quantifiable values, in which case it will be omitted.

If there are values above the BLQ, but too sparse to allow full analysis, descriptive statistics will be performed on available values.

#### 11.4.4.2 Pharmacodynamic/Activity Data

The evaluation of PD biomarkers will be based on absolute and percent change from baseline in serum levels of total IgG, IgG subtypes (IgG1-4), immunoglobulin A (IgA), immunoglobulin M (IgM), albumin, and CIC that will be summarized by cohort and timepoint.

### 11.4.4.3 Immunogenicity Data

Immunogenicity results will be summarized by cohort and timepoint. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

#### 11.4.4.4 PDAI Data

PDAI results will be summarized by score (total activity score, total damage score), cohort, and timepoint. Descriptive statistics will include absolute change from baseline, and percent change from baseline. PDAI will also be summarized by disease severity category, mild (0 to 8), moderate (9 to 24), and severe (≥25).

# 11.4.5 Analysis of Exploratory Endpoints

### 11.4.5.1 Corticosteroid Use

The evaluation of corticosteroid use during the study will be summarized by cohort and timepoint.

#### 11.4.5.2 Health-Related Quality of Life Data

HR-QoL results from the ABQoL and Skindex-29 assessments will be summarized by cohort and timepoint

# 11.4.5.3 Photography

The qualitative assessment of changes in appearance of skin and mucosal lesions as determined by photography presented by cohort and timepoint.

# 11.5 Interim Analysis

No interim analysis is planned.
## 12. STUDY MANAGEMENT

### 12.1 Regulatory and Ethical Considerations

### 12.1.1 Ethical Conduct

The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH E6 Tripartite Guideline (January 1997), and in general, be conducted in a manner consistent with the principles described in the Declaration of Helsinki. The Investigator will ensure that the conduct of the study complies with the basic principles of GCP as outlined in the current version of 21 CFR, subpart D, Part 312, "Responsibilities of Sponsors and Investigators", Part 50, "Protection of Human Subjects", and Part 56, "Institutional Review Boards".

### 12.1.2 Informed Consent

A signed informed consent form (ICF) in compliance with 21 CFR, Part 50.25(a) and Part 50.25(b) and the ICH guidelines, will be obtained from each subject before the subject is entered into the study and before any study screening procedure is performed that involves risk. The method of obtaining and documenting the informed consent will comply with ICH GCP and all applicable laws and regulations and will be subject to approval by the Sponsor.

The Investigator, or designee, is responsible for obtaining written informed consent from each subject (or the subject's legally authorized representative) participating in this study after a thorough and clear explanation of the objectives, procedures, anticipated benefits, and potential hazards of the study. In the case where the subject is unable to read, an impartial witness should be present during the entire informed consent discussion. After the subject has orally consented to participation in the trial, the witness' signature on the form will attest that the information in the consent form was accurately explained and understood. The study site must retain the original ICF and a copy must be provided to the subject or to the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

The Sponsor, or designee, must review the signed ICF against any proposed deviations from a sample ICF the Sponsor has supplied to each site. The final IRB-approved document must be provided to the Sponsor for regulatory purposes.

The eCRF for this study contains a section for documenting informed subject consent, and this must be completed appropriately. Signed ICFs must remain in each subject's study file and must be available for verification by site monitors at any time. If new safety information results in significant changes in the risk/benefit assessment, the consent form should be reviewed and updated as necessary. All subjects (including those already being treated) should be informed of the new information, should be given a copy of the revised form, and should give their consent to continue in the study.

### 12.1.3 Subject Confidentiality and Privacy

As applicable, in accordance with the Health Insurance Portability and Accountability Act (HIPAA), and associated privacy regulations, a patient authorization to use personally

identifiable health information may be required from each patient before research activities begin.

The Investigator must ensure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On eCRFs or other documents submitted to the Sponsor, subjects should be identified by an identification code and not by their names. The Investigator should keep a subject enrollment log showing codes, names, and addresses. The Investigator should maintain documents intended for storing onsite (eg, subjects' written consent forms) in strict confidence.

All study drugs, subject bodily fluids and tissue, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by the Sponsor.

### 12.1.4 Future Use of Stored Specimens

Not all the tissue and blood components obtained during this study may be required for the tests that are part of the clinical trial. Available samples may be used for additional research. This research will help to understand disease subtypes, drug response, and AEs, and possibly identify new drug targets or biomarkers that predict subject response to treatment. The use of the samples for internal research will adhere to the guidelines defined by the FDA in "Guidance on Informed Consent for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individual Identifiable" (issued 25 April 2006) and the European Medicines Agency (EMA) "Reflection Paper on Pharmacogenetic Samples, Testing and Data Handling" (Doc. Ref. EMEA/CHMP/PGxWP/201914/2006; 15 November 2007). If a subject requests destruction of their tissue and blood samples and the samples have not yet been de-identified, the Sponsor will destroy the samples as described in the FDA guidance. The Sponsor will notify the Investigator in writing that the samples have been destroyed.

### 12.2 Study Administration

The study administration structure is provided in Table 10.





# 12.2.1 Institutional Review Board Approval

This study is being conducted under US IND 132727. This protocol (and any modifications) and appropriate consent procedures must be reviewed and approved by the site-specific IRB before the study is initiated. The IRB must operate in accordance with the current federal or local regulations. The Investigator will send a letter or certificate of IRB approval to the Sponsor (or designee) before subject enrollment and whenever subsequent modifications to the protocol are made.

### 12.2.2 Data Handling and Record Keeping

All data will be entered in a validated electronic data capture system using single data entry. Standard procedures (including following data review guidelines, manual clinical review based on subject profiles, computerized validation to produce queries, and maintenance of an audit file, which includes all database modifications) will be followed to ensure accurate data. Clinical personnel will review all data listings for outliers, data inconsistencies, and spelling errors.

### 12.2.3 Data Protection

The Investigator agrees that all information received from the Sponsor, including but not limited to the IB, this protocol, eCRFs, the INDs, and any other study information remain the sole and exclusive property of the Sponsor during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) or otherwise into the public domain without prior written consent from the Sponsor.

### 12.2.4 Study Site Regulatory Documentation

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should

be classified into 2 separate categories as follows: (1) Investigator's study file and (2) subject clinical source documents (see Section 12.2.5).

The Investigator's study file will contain the protocol and protocol amendments, eCRFs, query forms, IRB and governmental approval with correspondence, sample informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

Subject clinical source documents (usually predefined by the project to record key efficacy and safety parameters independent of the eCRFs) may include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, electroencephalogram, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject screening and enrollment logs. The Investigator must keep these two categories of documents on file for at least 2 years following the marketing application approval date for the study treatment and for the indication being investigated or for 2 years after the development program is discontinued and the FDA notified. After that period, the documents may be destroyed subject to local regulations with prior written permission from the Sponsor. If the Investigator wants to assign the study records to another party or move them to another location, the Sponsor must be notified in advance.

If the Investigator cannot guarantee the archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and the Sponsor to store these in a sealed container outside of the study site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storing outside of the study site.

### 12.2.5 Subject Clinical Source Documents and Background Data

Investigators must maintain adequate and accurate source documents on which the eCRFs for each subject are based. They are separate and distinct from the eCRFs.

These records include detailed notes on the following:

- Medical history
- Informed consent
- HIPAA authorization, if applicable (either contained in the ICF or presented to the subject candidate as a standalone document)
- Description of the complete consenting process
- The basic identifying information that linked the subject's medical record with the eCRFs
- The results of all diagnostic tests performed, diagnoses made, therapy provided, and any other data on the condition of the subject
- The medical condition of the subject during their involvement in the study
- All AEs
- The subject's exposure to the study medication
- The subject's exposure to any concomitant therapy
- All relevant observations and data on the condition of the subject throughout the trial
- Justification for all entries in the subject's eCRF

A subject log of all potentially eligible subjects considered, but not consented, for obvious deviations from the entry criteria, will be kept at each site. The log will contain subjects' initials, diagnosis, eligibility, or, if not eligible, reason for not consenting. All consented subjects will be logged, regardless of whether they ultimately enroll.

Upon request, the Investigator will supply the Sponsor with any required background data from the study documentation or clinic records. This is particularly important when eCRFs are illegible or when errors in data transcription are suspected. In case of special problems or governmental queries or requests for audit inspections, it is also necessary to have access to the complete study records, provided that subject confidentiality is protected.

### 12.2.6 Electronic Case Report Forms

Clinical trial data for this study will be captured on eCRF designed for computer processing and analysis. This computerized system will be validated and compliant with 21 CFR Part 11, as described in the FDA guidance "Use of Electronic Records and Electronic Signatures in Clinical Investigations Under 21 CFR Part 11 – Questions and Answers." If corrections are made after review and sign-off by the Investigator, he/she must be aware of the changes and provide written acknowledgement. There will also be an electronic audit trail. Corrections on paper CRFs must be initialed and dated by the person making the change. The Investigator agrees to provide all information requested on the eCRF in an accurate manner using instructions provided. The Investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported to Syntimmune in the eCRF and in all required reports.

An eCRF is required to be submitted for every subject who receives any amount of study drug. This includes submission of retrievable data on subjects who withdraw before completion of the study. Prior to submission, eCRFs must be reviewed for completeness and accuracy, and signed and dated where indicated, by the Investigator or designee. If a subject stops treatment or terminates from the study, the dates and reasons must be noted on the eCRF.

# 12.3 Clinical Monitoring, Audits, and Inspections

The Investigator and study staff are responsible for maintaining a comprehensive and accurate filing system of all study-related documentation that will be suitable for inspection for routine monitoring, audit, or inspection at any time by the Sponsor (or designee) and/or a regulatory authority.

### 12.3.1 Clinical Monitoring

During the clinical study, it is understood that the responsible Sponsor site monitor or designee (eg, contract research organization [CRO]) will contact and visit the study site at regular intervals for routine monitoring of various records. Routine monitoring activities will be conducted to verify adherence to the protocol, completeness, consistency and accuracy of the data, and to review study source documents and drug accountability records. Regular review of the eCRFs for completeness, clarity, and to cross-check against source documents is required to

 Syntimmune, Inc.

monitor the progress of the study. Data will be reviewed and verified against the source documents (eg, original medical records and laboratory results) to ensure validity.

The Investigator will provide the Sponsor or designee with full access to all source data (including laboratory tests) and provide administrative support if requested. The Investigator (or designee) must agree to cooperate with the site monitor to ensure that any problems detected during these monitoring visits are resolved.

Site-specific study procedures, such data-recording and handling of the data, may be assessed during the study by a Clinical Quality Assurance representative(s) authorized by the Sponsor. Further, this designee, as well as the site monitor, will be permitted to inspect the study documents (study protocol, eCRFs, study drug accountability, original study-relevant medical records) to ensure that the study is conducted in compliance with the protocol.

During these visits, all representatives of the Sponsor will be responsible for ensuring data integrity and subject confidentiality is protected.

### 12.3.2 Audits and Inspections

Clinical site and study audits will be conducted as necessary to assure the validity of the study data. The Sponsor (or designee) may perform a quality assurance audit to ensure compliance with GCP, this protocol, and all applicable regulatory requirements. The Investigator should ensure that study documents (protocol, eCRFs, study drug record-keeping, original study-relevant medical records) are made available to the Sponsor (or designee) for examination. All subject data will be treated as confidential.

A regulatory authority, after appropriate notification, may also wish to conduct an inspection during the study or even after its completion. If a regulatory authority requests an inspection, the Investigator must immediately inform the Sponsor.

### 12.4 Changes to the Protocol

Protocol modifications to ongoing studies must be made only after consultation between a Sponsor representative and the Investigator. Protocol modifications will be prepared, reviewed, and approved by Sponsor representatives.

All protocol modifications must be submitted to the IRB for information and approval in accordance with local requirements, and to regulatory agencies, if required. Approval must be obtained before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to study subjects, or when the change involves only logistical or administrative aspects of the trial (eg, change in site monitor, change of telephone number).

### 12.5 Study Discontinuation and Closure

The Sponsor has the right to terminate the study at any time. In terminating the study, the Sponsor and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests.

# 13. PUBLICATION AND DATA SHARING POLICY

The results of this study may be published or presented at scientific meetings. The Investigator agrees that any manuscript or abstract they author may be published only after receiving written permission from the Sponsor.

If the Sponsor coordinates a publication or presentation of study results from all study sites, the participation of Investigator or other representatives of study site as a named author shall be determined in accordance with the Sponsor's policy and generally accepted standards for authorship as developed by the International Committee of Medical Journal Editors (ICMJE) and in accordance with Good Publication Practices.

### 14. REFERENCES

Agarwal S, Cunningham-Rundles C. Assessment and clinical interpretation of reduced IgG values. Ann Allergy Asthma Immunol. 2007;99(3):281-3.

Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID), which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. Clin Exp Immunol. 2013;174(2):203-11.

Blaha M, Pitha J, Blaha V, Lanska M, Maly J, Filip S, et al. Experience with extracorporeal elimination therapy in myasthenia gravis. Transfus Apher Sci. 2011;45(3):251-6.

Chren MM, Lasek RJ, Quinn LM, Mostow EN, Zyzanski SJ. Skindex, a quality-of-life measure for patients with skin disease: reliability, validity, and responsiveness. J Invest Dermatol. 1996;107(5):707-13.

Eming R, Hertl M. Immunoadsorption in pemphigus. Autoimmunity. 2006;39(7):609-16.

Furst DE. Serum immunoglobulins and risk of infection: how low can you go? Semin Arthritis Rheum. 2009;39(1):18-29.

Gonzalez-Quintela A, Alende R, Gude F, Campos J, Rey J, Meijide LM, et al. Serum levels of immunoglobulins (IgG, IgA, IgM) in a general adult population and their relationship with alcohol consumption, smoking and common metabolic abnormalities. Clin Exp Immunol. 2008;151(1):42-50.

Hsu DY, Brieva J, Sinha AA, Langan SM, Silverberg JI. Comorbidities and inpatient mortality for pemphigus in the U.S.A. Br J Dermatol. 2016;174(6):1290-8.

Jolliff CR, Cost KM, Stivrins PC, Grossman PP, Nolte CR, Franco SM, et al. Reference intervals for serum IgG, IgA, IgM, C3, and C4 as determined by rate nephelometry. Clin Chem. 1982;28(1):126-8.

Kasperkiewicz M, Ellebrecht CT, Takahashi H, Yamagami J, Zillikens D, Payne AS, et al. Pemphigus. Nat Rev Dis Primers. 2017;3:17026.

Keystone E, Fleischmann R, Emery P, Furst DE, van Vollenhoven R, Bathon J, et al. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007;56(12):3896-908.

Kohler W, Bucka C, Klingel R. A randomized and controlled study comparing immunoadsorption and plasma exchange in myasthenic crisis. J Clin Apher. 2011;26(6):347-55.

Langan SM, Smeeth L, Hubbard R, Fleming KM, Smith CJ, West J. Bullous pemphigoid and pemphigus vulgaris--incidence and mortality in the UK: population based cohort study. BMJ. 2008;337:a180.

McMillan SA, Douglas JP, Archbold GP, McCrum EE, Evans AE. Effect of low to moderate levels of smoking and alcohol consumption on serum immunoglobulin concentrations. J Clin Pathol. 1997;50(10):819-22.

Nixon AE, Chen J, Sexton DJ, Muruganandam A, Bitonti AJ, Dumont J, et al. Fully human monoclonal antibody inhibitors of the neonatal fc receptor reduce circulating IgG in non-human primates. Front Immunol. 2015;6:176.

Roopenian DC, Christianson GJ, Sproule TJ, Brown AC, Akilesh S, Jung N, et al. The MHC class I-like IgG receptor controls perinatal IgG transport, IgG homeostasis, and fate of IgG-Fc-coupled drugs. J Immunol. 2003;170(7):3528-33.

Rosenbach M, Murrell DF, Bystryn JC, Dulay S, Dick S, Fakharzadeh S, et al. Reliability and convergent validity of two outcome instruments for pemphigus. J Invest Dermatol. 2009;129(10):2404-10.

Schmaldienst S, Mullner M, Goldammer A, Spitzauer S, Banyai S, Horl WH, et al. Intravenous immunoglobulin application following immunoadsorption: benefit or risk in patients with autoimmune diseases? Rheumatology. 2001;40(5):513-21.

Sebaratnam DF, Hanna AM, Chee SN, Frew JW, Venugopal SS, Daniel BS, et al. Development of a quality-of-life instrument for autoimmune bullous disease: the Autoimmune Bullous Disease Quality of Life questionnaire. JAMA Dermatol. 2013;149(10):1186-91.

Sebaratnam DF, Okawa J, Payne A, Murrell DF, Werth VP. Reliability of the autoimmune bullous disease quality of life (ABQOL) questionnaire in the USA. Qual Life Res. 2015;24(9):2257-60.

Shimizu T, Takebayashi T, Sato Y, Niizeki H, Aoyama Y, Kitajima Y, et al. Grading criteria for disease severity by pemphigus disease area index. J Dermatol. 2014;41(11):969-73.

van Vollenhoven RF, Emery P, Bingham CO, 3rd, Keystone EC, Fleischmann RM, Furst DE, et al. Long-term safety of rituximab in rheumatoid arthritis: 9.5-year follow-up of the global clinical trial programme with a focus on adverse events of interest in RA patients. Ann Rheum Dis. 2013;72(9):1496-502.

# APPENDIX 1. NCI CTCAE, VERSION 4.03

 Syntimmune, Inc.

# Common Terminology Criteria for Adverse Events (CTCAE)

# Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

### Common Terminology Criteria for Adverse Events v4.0 (CTCAE)

### Quick Reference

The NCI Common Terminology Criteria Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

### **Components and Organization**

### SOC

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e. SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

### **CTCAE Terms**

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disea temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analysis Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

# Publish Date: May 28, 2009

# Definitions

A brief definition is provided to clarify the meaning of each AE term.

### Grades

displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic telephone, managing money, etc. observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; medications, and not bedridden. limiting age-appropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than e options for Grade selection.

Grade refers to the severity of the AE. The CTCAE Grade 5 (Death) is not appropriate for some AEs displays Grades 1 through 5 with unique clinical and therefore is not an option.

### ctivities of Daily Living (ADL)

- Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the
- Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking

<sup>†</sup> CTCAE v4.0 incorporates certain elements of the MeduRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).

### CONTENTS

| SOC | Page |
|---------------------------------------------------------------------|------|
| Blood and lymphatic system disorders | 3 |
| Cardiac disorders | 4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 9 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | 76 |
| Vascular disorders | 77 |

| | В | lood and lymphatic system | em disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 2 | | 3 | 4 | 5 |
| Anemia | Hemoglobin (Hgb) <lln -="" 10.0<br="">g/dL; <lln -="" -<br="" 6.2="" <lln="" l;="" mmol="">100 g/L</lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L;<br><80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an reduction in the amount of palpitations of the heart, soft syst | • | • • • | ay include pallor of the skin and m | ucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25% reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50% reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder characteriz | ed by the inability of the bone mar | row to produce hematopoietic ele | ments. | | |
| Disseminated intravascular<br>coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by systemic pathological activa<br>s depleted of platelets and coagula | - | which results in clot formation thro | oughout the body. There is an incr | ease in the |
| Febrile neutropenia | - | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>degrees F) for more than one ho | ed by an ANC <1000/mm3 and a sur. | single temperature of >38.3 degre | es C (101 degrees F) or a sustain | ed temperature of >=38 degrees 0 | (100.4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate widespread erythrocyte ce | Il membrane destruction. | I | 1 |
| Hemolytic uremic syndrome | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteriz | ed by a form of thrombotic microa | ngiopathy with renal failure, hemo | lytic anemia, and severe thromboo | ytopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of leucostasis; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate an increased number of w | nite blood cells in the blood. | | |
| _ymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in a lymph node. | | | |
| Spleen disorder | Incidental findings (e.g., Howell-<br>Jolly bodies); mild degree of<br>thrombocytosis and<br>leukocytosis | Prophylactic antibiotics indicated | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder of the splee | en. | | , | | |
| Thrombotic thrombocytopenic purpura | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | iled by the presence of microangion<br>all disturbances. It is an acute or s | • | r<br>cytopenic purpura, fever, renal abr | ' | malities suc |
| Blood and lymphatic system | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| disorders - Other, specify | symptomac or finid<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | noninvasive intervention indicated; limiting age-appropriate instrumental ADL | but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | urgent intervention indicated | Deall |

| Cardiac disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute coronary syndrome | - | Symptomatic, progressive angina; cardiac enzymes normal; hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | | • | dium secondary to coronary artery | disease. The clinical presentation | covers a |
| | unstable angina to myocardial infa | | | Life ii | L |
| Aortic valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in aortic valve func | tion or structure. | I | T | |
| Asystole | Periods of asystole; non-urgent medical management indicated | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia without cardi | ac electrical activity. Typically, this | is accompanied by cessation of the | ne pumping function of the heart. | |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>originates above the ventricles. | ed by a dysrhythmia without disce | rnible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz atria. | ed by a dysrhythmia with organize | ed rhythmic atrial contractions with | a rate of 200-300 beats per minut | e. The rhythm disturbance origina | tes in the |
| Atrioventricular block complete | - | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with complet | e failure of atrial electrical impulse | conduction through the AV node t | o the ventricles. | |
| Atrioventricular block first<br>degree | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | - | - | - |
| | ed by a dysrhythmia with a delay interval greater than 200 milliseco | • | ction of an electrical impulse throug | th the atrioventricular (AV) node be | eyond 0. |
| Cardiac arrest | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by cessation of the pumping fu | nction of the heart. | | | |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by substernal discomfort due to | o insufficient myocardial oxygenati | ion. | | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by pathological irregularities in | the cardiac conduction system. | | | |
| Constrictive pericarditis | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | 1 | cardial sact these fibrotic changes | i mpede normal myocardial function | 1 | e action. |
| Definition: A disorder characteriz | ed by a thickened and fibrotic peri | odraidi odo, triodo librotio oridrigos | | | |

| | | Cardiac disorde | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic | - | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | ed by failure of the left ventricle to ea, orthopnea, and other signs ar | | e an increase in distending pressure stion and edema. | e and in end-diastolic volume. Clin | ical |
| Mitral valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characterize | ed by a defect in mitral valve funct | tion or structure. | | T | |
| Mobitz (type) II atrioventricular<br>olock | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with relatively<br>trioventricular (AV) node to the ve | · | block of an atrial impulse. This is t | he result of intermittent failure of a | trial electi |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a progre<br>n through the atrioventricular (AV | | ior to the blocking of an atrial impu | llse. This is the result of intermitter | nt failure o |
| Myocardial infarction | - | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences;<br>hemodynamically unstable | Death |
| Definition: A disorder characterize | ed by gross necrosis of the myoca | ardium; this is due to an interruption | on of blood supply to the area. | | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characterize | ed by inflammation of the muscle | tissue of the heart. | | | |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | - | - | - |
| Definition: A disorder characterize | ed by an unpleasant sensation of | irregular and/or forceful beating o | f the heart. | <b>.</b> | |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characterize originates in the atria. | ed by a dysrhythmia with abrupt o | nset and sudden termination of at | rial contractions with a rate of 150- | -250 beats per minute. The rhythm | disturba |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by fluid collection within the pe | ricardial sac, usually due to inflam | mation. | | |
| Pericardial tamponade | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an increase in intrapericardi | al pressure due to the collection of | of blood or fluid in the pericardium. | | |
| Pericarditis | Asymptomatic, ECG or physical findings (e.g., rub) consistent | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic consequences (e.g., pericardial | Life-threatening consequences; urgent intervention indicated | Death |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe<br>regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in pulmonary valve | function or structure. | <u> </u> | 1 | , |
| Restrictive cardiomyopathy | - | - | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | ed by an inability of the ventricles | | | | I |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., ventricular assist device);<br>heart transplant indicated | Death |
| Definition: A disorder characteriz | ed by impairment of right ventricul | ar function associated with low eje | ection fraction and a decrease in n | notility of the right ventricular wall. | |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with alternation | | 1 | | 1 |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical intervention indicated | Severe, medically significant, medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | | that originates in the sinus node. | | |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates in the sinus no | ode. | 1 |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per min | nute that originates above the ven | tricles. | |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| | ed by a defect in tricuspid valve fu | | | | |
| Ventricular arrhythmia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia that originate | s in the ventricles. | Ι | 1 | |
| Ventricular fibrillation | - | - | - | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz ventricles. | ed by a dysrhythmia without disce | rnible QRS complexes due to rapi | d repetitive excitation of myocardi | al fibers without coordinated contr | action of the |
| Ventricular tachycardia | - | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates distal to the bu | undle of His. | |
| Wolff-Parkinson-White syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of an accessor | ry conductive pathway between th | e atria and the ventricles that caus | ses premature ventricular activatio | n. |
| Cardiac disorders - Other,<br>specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Congenital, familial and genetic disorders | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Congenital, familial and genetic disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Ear and labyrinth dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the ear. | | | |
| External ear inflammation | External otitis with erythema or dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis; stenosis or osteomyelitis; necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation, swelling and r | edness to the outer ear and ear c | anal. | | |
| External ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the external ear region. | · | <b>.</b> | |
| Hearing impaired | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: subjective change in hearing in the absence of documented hearing loss. Pediatric (on a 1, 2, 3, 4, 6 and | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated. Adults not enrolled in Monitoring Program: hearing loss with hearing aid or intervention indicated; limiting self care ADL. | Adults: Decrease in hearing to profound bilateral loss (absolute threshold >80 dB HL at 2 kHz and above); non-servicable hearing. Pediatric: Audiologic indication for cochlear implant and additional speech-language related services indicated. | - |
| | 8 kHz audiogram): Threshold<br>shift >20 dB at 8 kHz in at least<br>one ear. | Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 4 kHz and above in at least one ear. | Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing aids; threshold shift >20 dB at 3 kHz and above in at least one ear; additional speech-language related services indicated. | | |
| | ted by partial or complete loss of th | | | | I |
| Middle ear inflammation | Serous otitis | Serous otitis, medical intervention indicated | Mastoiditis; necrosis of canal soft tissue or bone | Life-threatening consequences; urgent intervention indicated | Death |
| | red by inflammation (physiologic re | i i | | | |
| Tinnitus | Mild symptoms; intervention not indicated | instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Vertigo | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz vertigo). | eed by a sensation as if the externa | 1 | ı | I<br>he himself were revolving in space | l<br>e (subjective |
| Vestibular disorder | - | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by dizziness, imbalance, nause | ea, and vision problems. | | | |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Endocrine disord | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adrenal insufficiency | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | irs when the adrenal cortex does not<br>lison's disease or primary adrenal in: | · - | cortisol and in some cases, the ho | ormone aldosterone. It may be due | to a disorde |
| Cushingoid | Mild symptoms; intervention not indicated | intervention indicated | Severe symptoms, medical intervention or hospitalization indicated | - | - |
| Definition: A disorder character<br>osteoporosis, usually due to ex | rized by signs and symptoms that re<br>cogenous corticosteroids. | semble Cushing's disease or synd | drome: buffalo hump obesity, striat | ions, adiposity, hypertension, diab | etes, and |
| Delayed puberty | - | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | - | - |
| Definition: A disorder character | rized by unusually late sexual maturi | ity. | ' | • | • |
| Growth accelerated | - | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | - | - |
| Definition: A disorder character | rized by greater growth than expecte | ed for age. | | 1 | |
| Hyperparathyroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character<br>the blood). | rized by an increase in production of | parathyroid hormone by the para | thyroid glands. This results in hypo | ercalcemia (abnormally high levels | of calcium i |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid suppression therapy indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by excessive levels of thyroid h | normone in the body. Common car | uses include an overactive thyroid | gland or thyroid hormone overdos | e. |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical intervention or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | • | • |
| Hypothyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by a decrease in production of | | and. | | |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical markers of puberty for females <8 years and males <9 years | - | - | - |
| Definition: A disorder character<br>9 for boys. | rized by unusually early developmen | nt of secondary sexual features; th | e onset of sexual maturation begi | ns usually before age 8 for girls an | d before age |
| Virilization | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | rized by inappropriate masculinizatio | on occurring in a female or prepub | ertal male. | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| llurred vision | Intervention not indicated | Symptomatic; limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | terized by visual perception of u | nclear or fuzzy images. | ı | I | I |
| Cataract | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; moderate decrease in visual acuity (20/40 or better) | Symptomatic with marked decrease in visual acuity (worse than 20/40 but better than 20/200); operative intervention indicated (e.g., cataract surgery) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charac<br>intreated. | terized by partial or complete op | eacity of the crystalline lens of o | one or both eyes. This results ir | n a decrease in visual acuity an | d eventual blindness if |
| Conjunctivitis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; topical intervention indicated (e.g., antibiotics); limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | terized by inflammation, swelling | and redness to the conjunctiv | a of the eye. | | |
| Corneal ulcer | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Limiting self care ADL;<br>declining vision (worse than<br>20/40 but better than 20/200) | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Definition: A disorder charac | terized by an area of epithelial ti | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the cornea | and anterior chamber. |
| Dry eye | Asymptomatic; clinical or diagnostic observations only; mild symptoms relieved by lubricants | Symptomatic; multiple<br>agents indicated; limiting<br>instrumental ADL | Decrease in visual acuity<br>(<20/40); limiting self care<br>ADL | - | - |
| Definition: A disorder charac | terized by dryness of the cornea | and conjunctiva. | | ' | • |
| Extraocular muscle paresis | Asymptomatic; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder charac | terized by incomplete paralysis | of an extraocular muscle. | ' | ' | ' |
| Eye pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder charac | terized by a sensation of marked | d discomfort in the eye. | | | |
| Eyelid function disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; nonoperative intervention indicated; limiting instrumental ADL | Limiting self care ADL;<br>operative intervention<br>indicated | - | - |
| Definition: A disorder charac | terized by impaired eyelid function | on.<br>I | I | Γ | |
| lashing lights | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charac | terized by a sudden or brief burs | st of light. | 1 | I | <b>I</b> |
| loaters | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| efinition: A disorder charac | terized by an individual seeing s | pots before their eyes. The sport | ots are shadows of opaque cell | fragments in the vitreous hume | or or lens. |
| Glaucoma | Elevated intraocular<br>pressure (EIOP) with single<br>topical agent for intervention;<br>no visual field deficit | EIOP causing early visual<br>field deficits; multiple topical<br>or oral agents indicated;<br>limiting instrumental ADL | EIOP causing marked visual<br>field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated;<br>limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charac | terized by an increase in pressu | re in the eyeball due to obstruc | ction of the aqueous humor out | flow. | |
| Ceratitis | - | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Decline in vision (worse than<br>20/40 but better than<br>20/200); limiting self care<br>ADL | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Antimitian, A diagrafar abaras | terized by inflammation to the co | ornea of the eye. | | | |
| Pelifilion. A disorder charac | 1 | | | | |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only | Limiting vision of the affected eye (20/40 or better) | eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| | erized by involvement of the op | 1 | ĺ | | 1 |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by swelling around the o | ptic disc.<br>T | <u> </u> | <u> </u> | |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charact | erized by fear and avoidance of | f light. | | | |
| Retinal detachment | Asymptomatic | Exudative and visual acuity<br>20/40 or better | Rhegmatogenous or<br>exudative detachment;<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by the separation of the | inner retina layers from the und | lerlying pigment epithelium. | | |
| Retinal tear | - | Laser therapy or pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by a small laceration of t | he retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | s and floaters. |
| Retinal vascular disorder | - | Topical medication indicated | Intravitreal medication; operative intervention indicated | - | - |
| Definition: A disorder charact | erized by pathological retinal bl | ood vessels that adversely affe | cts vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked<br>decrease in visual acuity<br>(worse than 20/40);<br>disabling; limiting self care<br>ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder involvin | g the retina. | | | | |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better) | Symptomatic, limiting self care ADL; marked decrease in visual acuity (worse than 20/40) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by involvement of the sc | lera of the eye. | T | T | 1 |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | • | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by inflammation to the uv | vea of the eye. | Ι | Ι | T. |
| Vitreous hemorrhage | Asymptomatic or mild symptoms; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by blood extravasation in | nto the vitreous humor. | T | T | T |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | - | - |
| Definition: A disorder of excess | ssive tearing in the eyes; it can | be caused by overproduction of | of tears or impaired drainage of | the tear duct. | |
| Eye disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Sight-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | - |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension Definition: A disorder characteriz | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| | | Madanta a la Raitia | 0 | | |
| Abdominal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the abdominal region. | T | | |
| Anal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an abnormal communication | between the opening in the anal | canal to the perianal skin. | Г | |
| Anal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the anal region | on. | T | | |
| Anal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the anus. | | | |
| Anal necrosis | - | - | TPN or hospitalization indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | ed by a necrotic process occurring | | | | 1 |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the anal region. | T | | |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the anal canal. | | | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the anal ca | nal. | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by accumulation of serous or h | emorrhagic fluid in the peritoneal | cavity. | | |
| Bloating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | - | - | - |
| Definition: A disorder characteriz | ed by subject-reported feeling of u | incomfortable fullness of the abdo | men. | | |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the cecum. | | | | |
| Cheilitis | Asymptomatic; clinical or diagnostic observations only; | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | - | - |
| | intervention not indicated | | | | |

| Gastrointestinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| Advance France | Grade 1 2 3 4 | | | | |
| Adverse Event | 1 | | | 4 | |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the colon. | | | | |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the large intestine and | another organ or anatomic site. | | |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the colon. | T | T | Γ | |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated rized by blockage of the normal flow | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | Tized by blockage of the normal flow | | | | D41- |
| Colonic perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by a rupture in the colonic wall. | | | | ı |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the colon. | ' | ' | |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the colon. | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with regular use of laxatives or enemas; limiting instrumental ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by irregular and infrequent or d | ifficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis<br>or periapical abscess or<br>resulting in tooth loss | - | - |
| Definition: A disorder characte | rized by the decay of a tooth, in whice | h it becomes softened, discolored | and/or porous. | | |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day over baseline; moderate increase in ostomy output compared to baseline | Increase of >=7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by frequent and watery bowel r | novements. | | | |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment orally; tube feeding or TPN indicated; unstimulated saliva <0.1 ml/min | - | - |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the duodenum and and | other organ or anatomic site. | | |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the duodenur | n. | | 1 | I |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective operative intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of stomach contents through the | duodenum. | | |
| Duodenal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a rupture in the duodenal w | all. | 1 | 1 | 1 |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the duodenum. | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the duoder | nal wall. | |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| Definition: A disorder characto<br>heartburn, nausea and vomiti | erized by an uncomfortable, often pai | nful feeling in the stomach, resulti | ing from impaired digestion. Sympt | oms include burning stomach, blo | ating, |
| Dysphagia | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely altered eating/swallowing; tube feeding or TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by difficulty in swallowing. | 1 | • | ' | • |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent abdominal pain; fever; ileus; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the small ar | nd large intestines. | | 1 | 1 |
| Enterovesical fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the urinary bladder and | d the intestine. | | |
| Esophageal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | n between the esophagus and an | other organ or anatomic site. | | |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor | Transfusion, radiologic, endoscopic, or elective | Life-threatening consequences; urgent intervention indicated | Death |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | g in the esophageal wall. | | | |
| Esophageal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by blockage of the normal flow | | | I | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the esophageal region. | | | |
| Esophageal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a rupture in the wall of the e | 1 | | | |
| Esophageal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the esophagus. | | · | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammate | ory and necrotic erosive lesion on | the mucosal surface of the esopha | geal wall. | |
| Esophageal varices<br>hemorrhage | - | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from esophageal v | rarices. | | | |
| Esophagitis Definition: A disorder characte | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered eating/swallowing; oral supplements indicated | Severely altered<br>eating/swallowing; tube feeding,<br>TPN or hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Fecal incontinence | Occasional use of pads required | | Severe symptoms; elective | _ | _ |
| | | | operative intervention indicated | | |
| | mized by inability to control the escap | | | | |
| Flatulence | Mild symptoms; intervention not indicated | psychosocial sequelae | ] | - | - |
| Definition: A disorder characte | rized by a state of excessive gas in | | | I | |
| Gastric fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | n between the stomach and anoth | er organ or anatomic site. | T | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the gastric wa | all. | | 1 | |
| Gastric necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | I. | I . | 1 | 1 | 1 |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | 1 | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a rupture in the stomach wa | | T | | I |
| Gastric stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a narrowing of the lumen of | the stomach. | | <b>.</b> | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a circumscribed, inflammato | ĺ | | | |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | rized by inflammation of the stomach | l. | 1 | T | |
| Gastroesophageal reflux<br>disease | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | rized by reflux of the gastric and/or d<br>y result in injury to the esophageal m | | | nd usually caused by incompetend | ce of the lov |
| Gastrointestinal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site. | |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the gastrointestinal region | n. | • | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to<br>maintain nutrition with dietary<br>and lifestyle modifications; may<br>need pharmacologic<br>intervention | Weight loss; refractory to medical intervention; unable to maintain nutrition orally | - | - |
| Definition: A disorder character | rized by an incomplete paralysis of th | re muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small into | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to aliment orally | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the gingival region. | 1 | T | |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by bleeding from the hemorrho | | 1 | I | |
| Hemorrhoids | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder character | rized by the presence of dilated vein | s in the rectum and surrounding a | rea. | | |
| leal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | between the ileum and another o | organ or anatomic site. | | |
| leal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by bleeding from the ileal wall. | • | • | • | |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| leal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteria | zed by blockage of the normal flow | of the intestinal contents in the ile | eum. | i | |
| leal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by a rupture in the ileal wall. | | | T | |
| leal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri: | zed by a narrowing of the lumen of | the ileum. | | T | 1 |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the ileum. | I | |
| lleus | -<br>zed by failure of the ileum to transp | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | led by failure of the flediff to trainsp | Medical intervention or minor | Transfusion radiologic | Life threatening consequences: | Death |
| ntra-abdominal hemorrhage | | cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri: | zed by bleeding in the abdominal c | avity. | | | |
| Jejunal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri: | '<br>zed by an abnormal communication | n between the jejunum and anoth | er organ or anatomic site. | | • |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri: | zed by bleeding from the jejunal wa | all. | , | ! | ' |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri: | zed by blockage of the normal flow | of the intestinal contents in the je | ejunum. | | |
| Jejunal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri: | ਾ<br>zed by a rupture in the jejunal wall. | 1 | ı | 1 | • |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | '<br>zed by a narrowing of the lumen of | the jejunum. | · | ·<br> | · |
| lejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri: | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the jejunun | 1. | |
| ip pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Lower gastrointestinal | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| hemorrhage | | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | | cauterization indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by bleeding from the lower gas | strointestinal tract (small intestine, | large intestine, and anus). | T | 1 |
| Malabsorption | - | Altered diet; oral intervention indicated | Inability to aliment adequately;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inadequate absorption of nu | trients in the small intestine. Sym | ptoms include abdominal marked | discomfort, bloating and diarrhea. | |
| Mucositis oral | Asymptomatic or mild | Moderate pain; not interfering | Severe pain; interfering with oral | Life-threatening consequences; | Death |
| | symptoms; intervention not | with oral intake; modified diet | intake | urgent intervention indicated | |
| | indicated | indicated | | | |
| Definition: A disorder characte | erized by inflammation of the oral mu | cosal. | | I | |
| Nausea | Loss of appetite without | Oral intake decreased without | Inadequate oral caloric or fluid | - | - |
| | alteration in eating habits | significant weight loss, | intake; tube feeding, TPN, or | | |
| | | dehydration or malnutrition | hospitalization indicated | | |
| | erized by a queasy sensation and/or t | | | | |
| Obstruction gastric | Asymptomatic; clinical or | Symptomatic; altered GI | Hospitalization indicated; | Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated | function; limiting instrumental ADL | elective operative intervention | urgent operative intervention indicated | |
| | intervention not indicated | ,,,,,,, | indicated; limiting self care ADL; disabling | maioatou | |
| Definition: A disorder characte | ।<br>erized by blockage of the normal flow | of the contents in the stomach | <del>-</del> | I | ı |
| Oral cavity fistula | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered GI function; | Life-threatening consequences; | Death |
| Oral Cavily listula | diagnostic observations only; | function | TPN or hospitalization indicated; | urgent intervention indicated | Dealii |
| | intervention not indicated | Turiotion | elective operative intervention | argone intorvention indicated | |
| | | | indicated | | |
| Definition: A disorder characte | erized by an abnormal communication | n between the oral cavity and ano | ther organ or anatomic site. | | |
| Oral dysesthesia | Mild discomfort; not interfering | Moderate pain; interfering with | Disabling pain; tube feeding or | - | _ |
| , | with oral intake | oral intake | TPN indicated | | |
| Definition: A disorder characte | rized by a burning or tingling sensati | on on the lips, tongue or entire mo | outh. | ' | |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| · • | , | intervention or minor | endoscopic, or elective | urgent intervention indicated | |
| | | cauterization indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by bleeding from the mouth. | | | | |
| Oral pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the mouth, tongue or lips | | | |
| Pancreatic duct stenosis | | | Severely altered GI function; | Life-threatening consequences; | D41- |
| | Asymptomatic; clinical or | Symptomatic; altered GI | Severely altered Griunction, | Life-tilleaterling consequences, | Death |
| | Asymptomatic; clinical or diagnostic observations only; | function | tube feeding or hospitalization | urgent operative intervention | Death |
| | | | tube feeding or hospitalization indicated; elective operative | | Death |
| | diagnostic observations only; | | tube feeding or hospitalization | urgent operative intervention | Death |
| Definition: A disorder characte | diagnostic observations only; | function | tube feeding or hospitalization indicated; elective operative | urgent operative intervention | Death |
| Definition: A disorder characte<br>Pancreatic fistula | diagnostic observations only; intervention not indicated | function | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; | urgent operative intervention indicated Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; | function the pancreatic duct. | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | |
| | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or | function the pancreatic duct. Symptomatic; altered GI | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; | urgent operative intervention indicated Life-threatening consequences; | |
| | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; | function the pancreatic duct. Symptomatic; altered GI | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | |
| Pancreatic fistula | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention | |
| Pancreatic fistula<br>Definition: A disorder characte | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated | Death |
| Pancreatic fistula<br>Definition: A disorder characte | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function between the pancreas and another moderate symptoms; medical | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; | |
| Pancreatic fistula<br>Definition: A disorder characte | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function between the pancreas and anoth Moderate symptoms; medical intervention or minor | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated ther organ or anatomic site. Transfusion, radiologic, endoscopic, or elective | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated | Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by an abnormal communication Mild; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function n between the pancreas and anot! Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; | Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage Definition: A disorder characte | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function n between the pancreas and anot! Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, endoscopic, or elective operative intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by an abnormal communication Mild; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function n between the pancreas and anot! Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, endoscopic, or elective operative intervention indicated Tube feeding or TPN indicated; | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage Definition: A disorder characte | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by an abnormal communication Mild; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function n between the pancreas and anot! Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, endoscopic, or elective operative intervention indicated Tube feeding or TPN indicated; radiologic, endoscopic, or | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage Definition: A disorder characte Pancreatic necrosis | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of diagnostic observations only; intervention not indicated erized by an abnormal communication Mild; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function between the pancreas and anotal Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, endoscopic, or elective operative intervention indicated Tube feeding or TPN indicated; | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage Definition: A disorder characte Pancreatic necrosis Definition: A disorder characte | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of Asymptomatic; clinical or diagnostic observations only; intervention not indicated erized by an abnormal communication Mild; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function between the pancreas and anot! Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, endoscopic, or elective operative intervention indicated Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent operative intervention indicated | Death Death |
| Pancreatic fistula Definition: A disorder characte Pancreatic hemorrhage Definition: A disorder characte Pancreatic necrosis | diagnostic observations only; intervention not indicated erized by a narrowing of the lumen of diagnostic observations only; intervention not indicated erized by an abnormal communication Mild; intervention not indicated | the pancreatic duct. Symptomatic; altered GI function between the pancreas and anotal Moderate symptoms; medical intervention or minor cauterization indicated | tube feeding or hospitalization indicated; elective operative intervention indicated Severely altered GI function; tube feeding or TPN or hospitalization indicated; elective operative intervention indicated her organ or anatomic site. Transfusion, radiologic, endoscopic, or elective operative intervention indicated Tube feeding or TPN indicated; radiologic, endoscopic, or | urgent operative intervention indicated Life-threatening consequences; urgent operative intervention indicated Life-threatening consequences; urgent intervention indicated | Death |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteri. | zed by inflammation of the pancrea | S. | 1 | | |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or<br>gingivitis; multiple sites of<br>bleeding on probing; moderate<br>bone loss | Spontaneous bleeding; severe bone loss with or without tooth loss; osteonecrosis of maxilla or mandible | - | - |
| Definition: A disorder in the ging | ival tissue around the teeth. | | | <del> </del> | |
| Peritoneal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteria | zed by a necrotic process occurring | in the peritoneum. | 1 | Г | ı |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by inflammation of the rectum. | | | | |
| Rectal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | between the rectum and another | r organ or anatomic site. | | |
| Rectal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the rectal wall | and discharged from the anus. | | | |
| Rectal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri: | zed by inflammation of the mucous | membrane of the rectum. | | | |
| Rectal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri: | zed by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | zed by blockage of the normal flow | of the intestinal contents in the re | ctum. | Γ | |
| Rectal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | zed by a sensation of marked disco | | | | |
| Rectal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | zed by a rupture in the rectal wall. | T | 1 | | |
| Rectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri. | zed by a narrowing of the lumen of | the rectum. | | | |
| Rectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function (e.g. altered dietary habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | T | Grade | Г | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Retroperitoneal hemorrhage | -<br>zed by bleeding from the retroperite | Self-limited; intervention indicated | Transfusion, medical, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Salivary duct inflammation | Slightly thickened saliva; slightly | | Acute salivary gland necrosis; | Life-threatening consequences; | Death |
| Sanvary duct illinariffication | altered taste (e.g., metallic) | markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | severe secretion-induced<br>symptoms (e.g., thick saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated;<br>limiting self care ADL; disabling | urgent intervention indicated | Dealii |
| Definition: A disorder characteriz | ed by inflammation of the salivary | duct. | | | |
| Salivary gland fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by an abnormal communication | between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe pain; interfering with oral<br>intake; tube feeding, TPN or<br>hospitalization indicated; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the intestinal contents. | | | |
| Small intestinal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by a rupture in the small intesti | ne wall. | 1 | <u> </u> | |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the small intestine. | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the small in | itestine. | |
| Stomach pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | red by a sensation of marked disco | omfort in the stomach. | | | |
| Tooth development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with oral surgery | Maldevelopment with impairment not surgically correctable; disabling | - | - |
| Definition: A disorder characteriz | red by a pathological process of the | e teeth occurring during tooth dev | elopment. | Γ | |
| Tooth discoloration | Surface stains | - | - | - | - |
| Definition: A disorder characteriz | red by a change in tooth hue or tint | t. | 1 | 1 | |
| Toothache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Typhlitis | - | - | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal signs | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the cecum. | | | | |
| Upper gastrointestinal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the upper gas | trointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | |
| Vomiting | 1 - 2 episodes (separated by 5 minutes) in 24 hrs | 3 - 5 episodes (separated by 5 minutes) in 24 hrs | >=6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the reflexive act of ejecting t | he contents of the stomach throug | gh the mouth. | • | |
| Gastrointestinal disorders -<br>Other, specify | , , , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold;<br>shivering; chattering of teeth | Moderate tremor of the entire body; narcotics indicated | Severe or prolonged, not responsive to narcotics | - | - |
| Definition: A disorder chara | cterized by a sensation of cold that ofte | n marks a physiologic response to | sweating after a fever. | | |
| Death neonatal | - | - | - | - | Death |
| Definition: A disorder chara | cterized by cessation of life occurring de | uring the first 28 days of life. | | | |
| Death NOS | - | - | - | - | Death |
| Definition: A cessation of life | e that cannot be attributed to a CTCAE | term associated with Grade 5. | | | |
| Edema face | Localized facial edema | Moderate localized facial edema; limiting instrumental ADL | Severe swelling; limiting self care ADL | - | - |
| Definition: A disorder chara | cterized by swelling due to excessive flu | uid accumulation in facial tissues. | | 1 | 1 |
| Edema limbs | 5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection | >10 - 30% inter-limb discrepancy in volume or circumference at point of greatest visible difference; readily apparent obscuration of anatomic architecture; obliteration of skin folds; readily apparent deviation from normal anatomic contour; limiting instrumental ADL | >30% inter-limb discrepancy in volume; gross deviation from normal anatomic contour; limiting self care ADL | - | - |
| Definition: A disorder chara | cterized by swelling due to excessive flu | uid accumulation in the upper or lo | ower extremities. | | |
| Edema trunk | Swelling or obscuration of<br>anatomic architecture on close<br>inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour; limiting<br>instrumental ADL | Gross deviation from normal anatomic contour; limiting self care ADL | - | - |
| Definition: A disorder chara | cterized by swelling due to excessive flu | uid accumulation in the trunk area | T | T | |
| Facial pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder chara | cterized by a sensation of marked disco | omfort in the face. | | | |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest;<br>limiting instrumental ADL | Fatigue not relieved by rest, limiting self care ADL | - | - |
| Definition: A disorder chara | cterized by a state of generalized weak | ness with a pronounced inability to | summon sufficient energy to acc | omplish daily activities. | |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>104.0 degrees F) for <=24 hrs | >40.0 degrees C (>104.0 degrees F) for >24 hrs | Death |
| Definition: A disorder chara | cterized by elevation of the body's temp | erature above the upper limit of n | ormal. | 1 | |
| Flu like symptoms | Mild flu-like symptoms present | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder chara cough. | cterized by a group of symptoms simila | r to those observed in patients wit | h the flu. It includes fever, chills, b | ody aches, malaise, loss of appet | ite and dry |
| Gait disturbance | Mild change in gait (e.g., wide-<br>based, limping or hobbling) | Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL | Disabling; limiting self care ADL | - | - |
| Definition: A disorder chara | cterized by walking difficulties. | 1 | 1 | 1 | • |
| Hypothermia | - | 35 - >32 degrees C; 95 - >89.6 degrees F | 32 - >28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C; 82.4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>hypotension, pulmonary edema,<br>acidemia, ventricular fibrillation) | |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Infusion related reaction | Mild transient reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; | Life-threatening consequences; urgent intervention indicated | Death |
| | | hrs | hospitalization indicated for clinical sequelae | | |
| Definition: A disorder characterize | zed by adverse reaction to the infus | sion of pharmacological or biologic | | T | 1 |
| Infusion site extravasation | - | Erythema with associated symptoms (e.g., edema, pain, induration, phlebitis) | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by leakage of a pharmacologic<br>sation and marked discomfort at the | • | nfusion site into the surrounding ti | ssue. Signs and symptoms includ | e indurati |
| Injection site reaction | Tenderness with or without associated symptoms (e.g., warmth, erythema, itching) | Pain; lipodystrophy; edema; phlebitis | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an intense adverse reaction | (usually immunologic) developing | at the site of an injection. | | |
| Irritability | Mild; easily consolable | Moderate; limiting instrumental ADL; increased attention indicated | Severe abnormal or excessive response; limiting self care ADL; inconsolable | - | - |
| Definition: A disorder characteriz condition. | zed by an abnormal responsivenes | s to stimuli or physiological arousa | al; may be in response to pain, frig | ht, a drug, an emotional situation | or a medi |
| Localized edema | Localized to dependent areas, no disability or functional | Moderate localized edema and intervention indicated; limiting | Severe localized edema and intervention indicated; limiting | - | - |
| | impairment | instrumental ADL | self care ADL | | |
| Definition: A disorder characterize | zed by swelling due to excessive flu | uid accumulation at a specific anal | tomic site. | | |
| Malaise | Uneasiness or lack of well being | Uneasiness or lack of well being; limiting instrumental ADL | - | - | - |
| Definition: A disorder characteriz | zed by a feeling of general discomf | ort or uneasiness, an out-of-sorts | feeling. | | |
| Multi-organ failure | - | - | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | Life-threatening consequences<br>(e.g., vasopressor dependent<br>and oliguric or anuric or<br>ischemic colitis or lactic<br>acidosis) | Death |
| Definition: A disorder characterize | zed by progressive deterioration of | the lungs, liver, kidney and clotting | g mechanisms. | | |
| Neck edema | Asymptomatic localized neck edema | Moderate neck edema; slight<br>obliteration of anatomic<br>landmarks; limiting instrumental<br>ADL | Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by swelling due to an accumula | ation of excessive fluid in the neck | | | |
| Non-cardiac chest pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by discomfort in the chest unre | lated to a heart disorder. | | | |
| Pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | zed by the sensation of marked disc | comfort, distress or agony. | ·<br>I | ·<br>I | |
| Sudden death NOS | - | - | - | - | Death |
| Definition: An unexpected cessa | tion of life that cannot be attributed | to a CTCAE term associated with | Grade 5. | Γ | |
| General disorders and administration site conditions - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age- | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or | Life-threatening consequences; urgent intervention indicated | Death |
| Caron, apoony | not indicated | appropriate instrumental ADL | prolongation of existing hospitalization indicated; | | |

| Hepatobiliary disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bile duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Severely altered GI function;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a narrowing of the lumen of | the bile duct. | 1 | | |
| Biliary fistula | - | Symptomatic and intervention not indicated | Severely altered GI function;<br>TPN indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | n between the bile ducts and anoth | ner organ or anatomic site. | | |
| Cholecystitis | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by inflammation involving the g | jallbladder. It may be associated w | vith the presence of gallstones. | • | • |
| Gallbladder fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Symptomatic or severely altered<br>GI function; TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by an abnormal communication | n between the gallbladder and and | other organ or anatomic site. | | |
| Gallbladder necrosis | - | - | - | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | rized by a necrotic process occurring | g in the gallbladder. | | | |
| Gallbladder obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; IV fluids indicated <24<br>hrs | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by blockage of the normal flow | | | T | I |
| Gallbladder pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by a sensation of marked disco | omfort in the gallbladder region. | | _ | |
| Gallbladder perforation | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by a rupture in the gallbladder | wall. | | | |
| Hepatic failure | - | - | Asterixis; mild encephalopathy; limiting self care ADL | Moderate to severe encephalopathy; coma; life-threatening consequences | Death |
| | rized by the inability of the liver to m | etabolize chemicals in the body. L | aboratory test results reveal abnor | mal plasma levels of ammonia, bi | ilirubin, lac |
| dehydrogenase, and alkaline p | | 0 | Townskins in the Control of the Cont | 1 15- 41 | D" |
| Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by bleeding from the liver. | | | l . | |
| Hepatic necrosis | - | - | - | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by a necrotic process occurring | g in the hepatic parenchyma. | | | |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by a sensation of marked disco | omfort in the liver region. | | | |
| Perforation bile duct | - | - | Radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| D 6 10 A P A A A | ized by a sustance in the well -fit | l<br>extrahepatic or intrahepatic bile du | | | I |

| | Hepatobiliary disorders | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| | | Grade | | | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 | | | | |
| Portal hypertension | - | Decreased portal vein flow | Reversal/retrograde portal vein flow; associated with varices and/or ascites | Life-threatening consequences; urgent intervention indicated | Death | | | | |
| Definition: A disorder characterize | ed by an increase in blood pressu | re in the portal venous system. | | | | | | | |
| Portal vein thrombosis | - | Intervention not indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death | | | | |
| Definition: A disorder characterize | ed by the formation of a thrombus | (blood clot) in the portal vein. | | | | | | | |
| Hepatobiliary disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death | | | | |
| | | | disabling; limiting self care ADL | | | | | | |
| | | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug fever <38 degrees C (<100.4 degrees F); intervention not indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an adverse local or general | response from exposure to an alle | | | |
| Anaphylaxis | - | - | Symptomatic bronchospasm, with or without urticaria; parenteral intervention indicated; allergy-related edema/angioedema; hypotension | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an acute inflammatory react<br>resents with breathing difficulty, di | • | | | ypersensitivi |
| Autoimmune disorder | | | | | Dooth |
| Autoimmune disorder | Asymptomatic; serologic or<br>other evidence of autoimmune<br>reaction, with normal organ<br>function; intervention not<br>indicated | Evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder resulting fr | om loss of function or tissue destru | iction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individe | ual to his ow |
| Cytokine release syndrome | Mild reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | following initial improvement;<br>hospitalization indicated for<br>clinical sequelae (e.g., renal<br>impairment, pulmonary<br>infiltrates) | Life-threatening consequences;<br>pressor or ventilatory support<br>indicated | Death |
| Definition: A disorder characterize | red by nausea, headache, tachyca | rdia, hypotension, rash, and shorti | ness of breath; it is caused by the | release of cytokines from the cells | |
| Serum sickness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash, urticaria, antihistamines indicated | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV<br>fluids indicated | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| | red by a delayed-type hypersensiti<br>e foreign antigen. Symptoms inclu | | | | |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the abdominal cavity. | | T | |
| Anorectal infection | Localized; local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | ving the anal area and the rectum. | IV antibiotic antifungal or | Life threatening consequences: | Death |
| Appendicitis | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Deam |
| | rized by acute inflammation to the | | 1 | | ъ " |
| Appendicitis perforated | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by acute inflammation to the viceal wall rupture causes the releas | vermiform appendix caused by a pa | athogenic agent with gangrenous o | changes resulting in the rupture of | the |
| Arteritis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving an artery. | | | |
| Biliary tract infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the biliary tract. | 1 | ı | ı |
| Bladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bladder. | | | |
| Bone infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | | T | | |
| Breast infection | - | Local infection with moderate<br>symptoms; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | Severe infection; axillary<br>adenitis; IV antibacterial,<br>antifungal, or antiviral<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | 1 | | T | L |
| Bronchial infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bronchi. | 1 | 1 | 1 |
| Catheter related infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process that | arises secondary to catheter use. | | | |
| Cecal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | ed by an infectious process involv | | , and the second | 7 | |
| Cervicitis infection | ed by an inicollous process involv | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Cervicius imecuon | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | Death |
| | | antifungal, or antiviral) | radiologic or operative | g | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the uterine cervix. | | | |
| Conjunctivitis infective | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| | | | intervention indicated | 1 | l |
| | ed by an infectious process involv | ring the conjunctiva. Clinical manifo | · · | | I |
| Corneal infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, antifungal, or antiviral) | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | |
| | | and and an animal | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the cornea. | 1 | 1 | • |
| Cranial nerve infection | - '- | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring a cranial nerve. | _ | | 1 |
| Device related infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | 1 | l |
| | ed by an infectious process involv | T | T | I | I |
| Duodenal infection | - | Moderate symptoms; medical | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., oral antibiotics) | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | |
| | | 4.142.54.55) | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the duodenum. | ' | • | • |
| Encephalitis infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | severe changes in mental | | |
| | | | status; self-limited seizure | | |
| | | | activity; focal neurologic | | |
| | | 1 | abnormalities | 1 | l |
| | ed by an infectious process involv | ring the brain tissue. | | I | I |
| Encephalomyelitis infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ।<br>ring the brain and spinal cord tissu | 1 | 1 | 1 |
| Endocarditis infective | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | 20001 |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| | Ų. | | | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the endocardial layer of the he | eart. | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the endocardial layer of the he | Systemic intervention or | Blindness (20/200 or worse) | T- |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Enterocolitis infectious | · | Passage of >3 unformed stools | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Lineroconus imectious | | per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal | antiviral intervention indicated; radiologic, endoscopic, or | urgent intervention indicated | Deali |
| | | pain | operative intervention indicated;<br>profuse watery diarrhea with<br>signs of hypovolemia; bloody | | |
| | | | diarrhea; fever; severe<br>abdominal pain; hospitalization<br>indicated | | |
| Definition: A disorder characteri | <br>zed by an infectious process involv | ing the small and large intestines | Indicated | | I |
| Esophageal infection | _ | Local intervention indicated | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Looping Gai milooton | | (e.g., oral antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | Dodan |
| | | | intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the esophagus. | T | | |
| Eye infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated; | |
| | | antifungal, or antiviral) | radiologic or operative intervention indicated | enucleation | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the eye. | T | Γ | 1 |
| Gallbladder infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic, endoscopic, or operative intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the gallbladder. | | | |
| Gum infection | Local therapy indicated (swish | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | and swallow) | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotic, antifungal, antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the gums. | T | | |
| Hepatic infection | - | - | IV antibiotic, antifungal, or antiviral intervention indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | radiologic or operative intervention indicated | urgent intervention indicated | |
| Definition: A disorder characteri | l<br>zed by an infectious process involv | I<br>ing the liver | Intervention indicated | l | I |
| Hepatitis viral | Asymptomatic, treatment not | - | Symptomatic liver dysfunction; | Decompensated liver function | Death |
| | indicated | | fibrosis by biopsy; compensated cirrhosis; reactivation of chronic hepatitis | (e.g., ascites, coagulopathy, encephalopathy, coma) | |
| Definition: A disorder characteri | ।<br>zed by a viral pathologic process ir | l<br>volving the liver parenchyma | Inopatito | Į. | 1 |
| Infective myositis | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| • | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| Definition: A disorder characteri | <br>zed by an infectious process involv | ing the skeletal muscles | intervention indicated | I | I |
| Joint infection | - | Localized; local intervention | Arthroscopic intervention | Life-threatening consequences; | Death |
| | | indicated; oral intervention | indicated (e.g., drainage) or | urgent intervention indicated | |
| | | indicated (e.g., antibiotic, | arthrotomy (e.g., open surgical | | |
| | | antifungal, antiviral); needle | drainage) | | |
| | | aspiration indicated (single or multiple) | | | |
| Definition: A disorder characteri | ।<br>zed by an infectious process involv | | ı | I | I |
| Kidney infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| • | | | antiviral intervention indicated; | urgent intervention indicated | 1 |
| | | | radiologic, endoscopic, or | | |
| | | | operative intervention indicated | | 1 |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| .aryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an inflammatory process ir | nvolving the larynx. | i | i | 1 |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characte | erized by an infectious process invol | ving the lips. | | | |
| Lung infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invol | ving the lungs. | Т | T | |
| Lymph gland infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invol | ving the lymph nodes. | Τ | 1 | |
| Mediastinal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invol | ving the mediastinum. | <u> </u> | | |
| Meningitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by acute inflammation of the r | neninges of the brain and/or spinal | cord. | ' | • |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invol | ving a mucosal surface. | | | |
| Nail infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characte | erized by an infectious process invol | ving the nail. | Τ | T | |
| Otitis externa | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by an infectious process invol<br>nptoms include fullness, itching, swe | • | • | ve water exposure (swimmer's ea | r infectior |
| Otitis media | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invol | ving the middle ear. | | | |
| Ovarian infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | 1 | 1 | | I . | I |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involv | ing the pancreas. | , | , | |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | rized by an eruption consisting of pa | | | | p, and upper |
| Paronychia | Nail fold edema or erythema; disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical intervention or IV antibiotics indicated; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by an infectious process involv | ing the soft tissues around the nai | l. | T | |
| Pelvic infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process involv | 1 | I | I | 1 |
| Penile infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involv | ing the penis. | | | |
| Periorbital infection | rized by an infectious process involv | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Peripheral nerve infection | nized by an injectious process involv | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, antifungal, or antiviral) | | urgent intervention indicated | Death |
| | rized by an infectious process involv | ing the peripheral nerves. | | | |
| Peritoneal infection | | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process involv | ing the peritoneum. | | Γ | |
| Pharyngitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the throat. | | | | |
| Phlebitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the vein. Clinical manifestation | s include erythema, marked disco | mfort, swelling, and induration alo | ng the course |
| of the infected vein. | I | I | I | Γ | |
| Pleural infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic, endoscopic, or operative intervention indicated | | |
| Definition: A disorder characteriz | l<br>ed by an infectious process involvi | l<br>ing the pleura | operative intervention introduced | l | l . |
| | _ | 1 | IV antibiotic antifungal or | Life-threatening consequences; | Death |
| Troduce infection | | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | Boati |
| | | antibiotic, antifungal, antiviral) | radiologic, endoscopic, or | | |
| | | | operative intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the prostate gland. | I | I | |
| Definition: A disorder characterized by an infectious process involving the pleura. Prostate infection - Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral intervention indicated (e.g., antibiotic, antifungal, antiviral intervention indicated (e.g., antibiotic, antifungal, antiviral intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by an infectious process involving the prostate gland. Rash pustular - Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by a circumscribed and elevated skin lesion filled with pus. Rhinitis infective - Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by an infectious process involving the nasal mucosal. Salivary gland infection - Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) Definition: A disorder characterized by an infectious process involving the salivary gland. Scrotal infection - Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by an infectious process involving the scrotum. Sepsis - Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by the presence of pathogenic microorganisms in the blood stream that cause a rapic local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by the presence of pathogenic microorganisms in the blood stream that cause a rapic local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) Definition: A disorder characterized by an infectious process involving the mucous membranes of the paranasal sinuess. Skin infection Localized, local intervention indicated (e.g., antifunantiviral) | IV antibiotic, antifungal, or | - | - | | |
| | | | antiviral intervention indicated; | | |
| | | antifungal, or antiviral) | | | |
| Definition: A disorder characteriz | ।<br>ed by a circumscribed and elevate | l<br>ed skin lesion filled with nus | | <u> </u> | I |
| | _ | · | _ | _ | _ |
| | | · | | | |
| | | antifungal, or antiviral) | | | |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the nasal mucosal. | | | |
| Salivary gland infection | - | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | , , | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotic, antifungal, antiviral) | | | |
| Definition: A disorder characterize | d by an infectious process involvi | ing the calivary gland | Intervention indicated | | l |
| | ed by all lillections process lilvolvi | T | IV antibiotic antifungal or | Life-threatening consequences; | Death |
| Scrotal infection | - | · · | antiviral intervention indicated; | urgent intervention indicated | Death |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involving | ing the scrotum. | <u> </u> | <u> </u> | 1 |
| Sepsis | - | - | - | Life-threatening consequences; | Death |
| | | | | urgent intervention indicated | |
| | ed by the presence of pathogenic | | | | |
| Sinusitis | - | · · | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | radiologic, endoscopic, or | urgent intervention indicated | |
| | | , , | operative intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the mucous membranes of the | paranasal sinuses. | | |
| Skin infection | Localized, local intervention | Oral intervention indicated (e.g., | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | indicated | antibiotic, antifungal, antiviral) | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| Definition: A disorder characteriz | <br> | ing the elip | Intervention indicated | | |
| Small intestine infection | ed by an infectious process involvi | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Small intestine intection | - | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | Deam |
| | | antibiotic, antifungal, antiviral) | radiologic or operative | 9 | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the small intestine. | | T | |
| Soft tissue infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characteriz | l<br>ed by an infectious process involvi | l<br>ing soft tissues | I | I | I |
| Splenic infection | - an iniconous process involvi | ing cont noodes. | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Spierno irriconori | | | antiviral intervention indicated; | urgent intervention indicated | Dean |
| | | | radiologic or operative | = | |
| | | | intervention indicated | | |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | zed by an infectious process involv | ing the spleen. | I | I | 1 |
| Stoma site infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing a stoma (surgically created op | ening on the surface of the body). | I | |
| Tooth infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing a tooth. | T | T | 1 |
| Tracheitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an infectious process involv | | | | |
| Upper respiratory infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the upper respiratory tract (nos | se, paranasal sinuses, pharynx, la | rynx, or trachea). | |
| Urethral infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the urethra. | T | T | |
| Urinary tract infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ,<br>ing the urinary tract, most commo | nly the bladder and the urethra. | | • |
| Uterine infection | | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the endometrium. It may exten | d to the myometrium and parame | trial tissues. | • |
| Vaginal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing the vagina. | 1 | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by an infectious process involv | ing the vulva. | | | |
| Wound infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by an infectious process involv | ing the wound. | T | 1 | 1 |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | , <b>,</b> | , poisoning and procedu | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention | Limiting instrumental ADL; | Limiting self care ADL; elective | - <del>-</del> | _ |
| | indicated | operative intervention indicated | surgery indicated | | |
| Definition: A finding of damage in<br>Affected leg and foot. | to the ankle joint characterized by a | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | y moving th |
| Aortic injury | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | | | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage | to the aorta. | 1 | | l | |
| Arterial injury | Asymptomatic diagnostic | Symptomatic (e.g., | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| , , | finding; intervention not indicated | claudication); repair or revision not indicated | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage | to an artery. | | | | |
| Biliary anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | | |
| Deficitions A finalism of locks | not indicated | | intervention indicated | indicated | l |
| | of bile due to breakdown of a biliary | | | | D4h |
| Bladder anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | of urine due to breakdown of a blad | dder anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | |
| Bruising | Localized or in a dependent area | Generalized | - | - | - |
| Definition: A finding of injury of t | he soft tissues or bone characteriz | ed by leakage of blood into surrou | nding tissues. | | 1 |
| Burn | Minimal symptoms; intervention not indicated | Medical intervention; minimal debridement indicated | Moderate to major debridement or reconstruction indicated | Life-threatening consequences | Death |
| • . | integrity to the anatomic site of an depends on the length and intensi | | * * | nicals, direct heat, electricity, flame | es and |
| Dermatitis radiation | Faint erythema or dry | Moderate to brisk erythema; | Moist desquamation in areas | Life-threatening consequences; | Death |
| Joinnaulo radiation | desquamation | patchy moist desquamation, | other than skin folds and | skin necrosis or ulceration of full | Boati |
| | | mostly confined to skin folds | creases; bleeding induced by | thickness dermis; spontaneous | |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin graft indicated | |
| Definition: A finding of cutaneou | <br> s inflammatory reaction occurring a | <br>as a result of exposure to biologica | I<br>Illy effective levels of ionizing radia | 19 | I |
| Esophageal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| _sopriageal anastomotic leak | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | ।<br>due to breakdown of an esophagea | l anastomosis (surgical connection | ।<br>n of two separate anatomic structu | res). | |
| Fall | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding of sudden n | novement downward, usually result | ting in injury. | , | | |
| Fallopian tube anastomotic leak | Asymptomatic; clinical or | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | |
| Definition: A finding of leakage of | due to breakdown of a fallopian tub | e anastomosis (surgical connectio | n of two separate anatomic structu | ıres). | |
| Fallopian tube perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture o | f the fallopian tube wall. | 1 | | | |
| Fracture | Asymptomatic; clinical or | Symptomatic but non-displaced; | Severe symptoms; displaced or | Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated | immobilization indicated | open wound with bone exposure; disabling; operative | urgent intervention indicated | |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage de | ue to breakdown of a gastric anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Gastrointestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage de | ue to breakdown of a gastrointesti | nal anastomosis (surgical connect | tion of two separate anatomic struc | ctures). | |
| Gastrointestinal stoma necrosis | - | Superficial necrosis; intervention not indicated | Severe symptoms;<br>hospitalization or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of a necrotic | process occurring in the gastroint | estinal tract stoma. | | | |
| Hip fracture | - | Hairline fracture; mild pain;<br>limiting instrumental ADL; non-<br>surgical intervention indicated | Severe pain; hospitalization or intervention indicated for pain control (e.g., traction); operative intervention indicated | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise | - |
| Definition: A finding of traumatic | injury to the hip in which the contir | nuity of either the femoral head, fe | moral neck, intertrochanteric or su | btrochanteric regions is broken. | |
| Injury to carotid artery | - | - | Severe symptoms; limiting self<br>care ADL (e.g., transient<br>cerebral ischemia); repair or<br>revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the carotid artery. | | | | |
| Injury to inferior vena cava | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the inferior vena cava. | T | I | <u> </u> | |
| Injury to jugular vein | - | - | Symptomatic limiting self care<br>ADL; disabling; repair or<br>revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the jugular vein. | 1 | 1 | <u> </u> | |
| Injury to superior vena cava | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic; repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | the superior vena cava. | | | | |
| Intestinal stoma leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | contents from an intestinal stoma | (surgically created opening on the | T | 1 15- 41 | D4h |
| Intestinal stoma obstruction | | Self-limited; intervention not indicated | Severe symptoms; IV fluids,<br>tube feeding, or TPN indicated<br>>=24 hrs; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of blockage of | of the normal flow of the contents | of the intestinal stoma. | 1 | <u> </u> | |
| Intestinal stoma site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood leak | age from the intestinal stoma. | ·<br> | · | · | |
| Intraoperative arterial injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | an artery during a surgical proce | dure. | | | |
| Intraoperative breast injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |

| | | , poisoning and proced | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | o the breast parenchyma during a | | • | <del>-</del> | |
| Intraoperative cardiac injury | - | - | Primary repair of injured organ/structure indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the heart during a surgical proce | edure. | | | |
| Intraoperative ear injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection of injured organ/structure indicated; disabling (e.g., impaired hearing; impaired balance) | Life-threatening consequences; urgent intervention indicated | Death |
| | o the ear during a surgical proced | | | | I |
| Intraoperative endocrine injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the endocrine gland during a sui | rgical procedure. | | | |
| Intraoperative gastrointestinal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the gastrointestinal system durin | g a surgical procedure. | | | |
| Intraoperative head and neck<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the head and neck during a surg | ical procedure. | | | |
| Intraoperative hemorrhage | - | - | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical proc | edure. | ı | ! | • |
| Intraoperative hepatobiliary injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the hepatic parenchyma and/or | biliary tract during a surgical pro | cedure. | | |
| Intraoperative musculoskeletal<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the musculoskeletal system duri | ng a surgical procedure. | | | |
| Intraoperative neurological injury | Primary repair of injured organ/structure indicated of the nervous system during a sur | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | | Ĭ | 0 11 " | | Б. " |
| Intraoperative ocular injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the eye during a surgical proced | ure. | | | |
| Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the kidney during a surgical prod | cedure. | ·<br> | · | |
| Intraoperative reproductive tract injury | | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| Injury, poisoning and procedural complications Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | the reproductive organs during a | | | · | |
| Intraoperative respiratory injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the respiratory system during a s | surgical procedure. | | | |
| Intraoperative skin injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the skin during a surgical proced | ure. | | | |
| Intraoperative splenic injury | the prices during a surgical president | Primary repair of injured organ/structure indicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the spleen during a surgical proc | | Complete resection or | Life threatening concernance | Dooth |
| Intraoperative urinary injury Definition: A finding of damage to | Primary repair of injured organ/structure indicated the urinary system during a surg | Partial resection of injured organ/structure indicated ical procedure. | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Intraoperative venous injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| muaoperauve venous injury | organ/structure indicated | organ/structure indicated | reconstruction of injured organ/structure indicated; disabling | urgent intervention indicated | Deali |
| Definition: A finding of damage to | a vein during a surgical procedu | re. | · | | |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | urine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| <u> </u> | · · | nastomosis (surgical connection o | T ' | Í | 1 |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | indicated | Death |
| | | anastomosis (surgical connection | | ľ | |
| Postoperative hemorrhage | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; radiologic, endoscopic, or operative intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ccurring after a surgical procedur | | Figure 4 and 5 70 f | I the share to the | D |
| Postoperative thoracic procedure complication | - | Extubated within 24 - 72 hrs postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A finding of a previous | ly undocumented problem that oc | curs after a thoracic procedure. | 1 | I | |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental | Severe symptoms; elective operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of protrusion | of the intestinal stoma (surgically | created opening on the surface of | the body) above the abdominal su | ırface. | |
| Prolapse of urostomy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective operative intervention or major stomal revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of displacem | ent of the urostomy. | | | | |
| Radiation recall reaction (dermatologic) | Faint erythema or dry desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| Definition: A finding of acute skin | inflammatory reaction caused by | drugs, especially chemotherapeut | ic agents, for weeks or months fol | owing radiotherapy. The inflamma | tory reaction |
| is confined to the previously irrad | liated skin and the symptoms disa | ppear after the removal of the pha | rmaceutical agent. | <u> </u> | , |
| Rectal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of a rectal anasto | omosis (surgical connection of two | separate anatomic structures). | | , |
| Seroma | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; simple aspiration indicated | Symptomatic, elective radiologic<br>or operative intervention<br>indicated | - | - |
| Definition: A finding of tumor-like | collection of serum in the tissues. | Т | T | | |
| Small intestinal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the si | nall bowel. | |
| Spermatic cord anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of a spermatic co | ord anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Spinal fracture | Mild back pain; nonprescription analgesics indicated | Moderate back pain;<br>prescription analgesics<br>indicated; limiting instrumental<br>ADL | Severe back pain;<br>hospitalization or intervention<br>indicated for pain control (e.g.,<br>vertebroplasty); limiting self care<br>ADL; disability | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise | Death |
| Definition: A finding of traumatic i | injury to the spine in which the cor | intinuity of a vertebral bone is broke | en. | ! | 1 |
| Stenosis of gastrointestinal stoma | - | Symptomatic; IV fluids indicated <24 hrs; manual dilation at bedside | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | of the gastrointestinal stoma (surg | gically created opening on the surf | ace of the body). | <del> </del> | , |
| Stomal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characterize gastroenterostomy procedure. | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on t | he jejunal mucosal surface close t | to the anastomosis site following a | ı |
| Tracheal hemorrhage | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| rracriear nemormage | clinical or diagnostic exam;<br>intervention not indicated | intervention indicated | indicated; radiologic or<br>endoscopic intervention<br>indicated | urgent intervention indicated | Death |
| Definition: A finding of bleeding fr | rom the trachea. | T | T | Г | 1 |
| Tracheal obstruction | Partial asymptomatic<br>obstruction on examination<br>(e.g., visual, radiologic or<br>endoscopic) | Symptomatic (e.g., noisy airway breathing), no respiratory distress; medical intervention indicated (e.g., steroids); limiting instrumental ADL | Stridor; radiologic or endoscopic intervention indicated (e.g., stent, laser); limiting self care ADL | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | 1 | • | • | • | • |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| racheostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood leal | kage from the tracheostomy site. | | | | |
| Jreteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a ureteral ana | stomosis (surgical connection of to | vo separate anatomic structures). | T | |
| Jrethral anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a urethral ana | stomosis (surgical connection of to | vo separate anatomic structures). | I | |
| Jrostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | of contents from a urostomy. | 1 | <u> </u> | | |
| Jrostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or endoscopic repair or stent placement indicated | Altered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | | | | |
| Jrostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding | from the urostomy site. | ı | ı | I | 1 |
| Jrostomy stenosis | - | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | g of the opening of a urostomy. | T. | · | | |
| Uterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a uterine anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a rupture in the uterine wall. | | 0 | 1 15- 41 | D41- |
| /aginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vaginal anas | stomosis (surgical connection of tw | o separate anatomic structures). | i - | |
| /as deferens anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vas deferens | s anastomosis (surgical connection | n of two separate anatomic structu | res). | |
| ascular access complication | - | Device dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including pulmonary embolism or life-threatening thrombus | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Venous injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated; disabling | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | a vein. | | | | |
| Wound complication | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound; local care indicated | Hernia without evidence of<br>strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by<br>operative intervention indicated | Hernia with evidence of<br>strangulation; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| · · · · · · | Incisional separation of <=25% | 1 | Fascial disruption or dehiscence | Life threatening concessions | Dooth |
| Wound dehiscence | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound with local care; asymptomatic hernia or symptomatic hernia without evidence of strangulation | Hascial disruption or deniscence without evisceration; primary wound closure or revision by operative intervention indicated | Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| Definition: A finding of separation | of the approximated margins of a | surgical wound. | T | Г | 1 |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of traumatic | injury to the wrist joint in which the | continuity of a wrist bone is broke | en. | | |
| Injury, poisoning and procedural complications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Investigations | <b>S</b> | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | y test result in which the partial th | | | possible indicator of coagulopat | hy, a prolonge |
| , , | may occur in a variety of disease | | | | |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | | 1 , | 1 | 1 |
| Alkaline phosphatase increased | 1 | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | · | · | | |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen. | _ |
| Blood antidiuretic hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of antidiuretic horm | one in the blood specimen. | | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is as | ssociated with jaundice. | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotropl | nin in a blood specimen. | | |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; | Symptomatic; medical intervention indicated; limiting instrumental ADI | Severe symptoms; limiting self care ADL | - | - |
| Definition A finding board on lab | intervention not indicated | instrumental ADL | | | I |
| | oratory test results that indicate a | 1 | ormone in a blood specimen. | | 1 |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ,<br>bnormal levels of prolactin hormor | ne in a blood specimen. | ' | • |
| Carbon monoxide diffusing capacity decreased | 3 - 5 units below LLN; for follow-<br>up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | 6 - 8 units below LLN; for follow-<br>up, an asymptomatic decrease<br>of >5 - 8 units (ml/min/mm Hg)<br>below the baseline value | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., >Grade 2 hypoxia or >Grade 2 or higher dyspnea) | - | - |
| Definition: A finding based on lun | g function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | ' | • |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| · | t which indicates increased levels | of cardiac troponin I in a biologica | 1 | | 1 |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test resul | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | | ·<br> |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | |
| Cholesterol high | >ULN - 300 mg/dL; >ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL; >10.34 -<br>12.92 mmol/L | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | oratory test results that indicate h | gher than normal levels of cholest | terol in a blood specimen. | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in levels of creatine pho | osphokinase in a blood specimen. | | |

| | | Investigations | <u> </u> | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of creatinine in a b | iological specimen. | | |
| Ejection fraction decreased | - | Resting ejection fraction (EF) 50 - 40%; 10 - 19% drop from baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline | Resting ejection fraction (EF) <20% | - |
| Definition: The percentage compo<br>contraction. | uted when the amount of blood eje | ected during a ventricular contracti | on of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected interval prolonged | | QTc 481 - 500 ms | QTc >= 501 ms on at least two<br>separate ECGs | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| | i i | bnormally long corrected QT inter | | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75% decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of fibrinogen i | n a blood specimen. | • | • |
| Forced expiratory volume<br>decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on tes | t results that indicate a relative de | crease in the fraction of the forced | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| - | | igher than normal levels of the enz<br>roup from a gamma glutamyl pept | | | IIIIa- |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of growth hormone | in a biological specimen. | • | |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of haptoglobir | in a blood specimen. | • | |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN | Increase in >4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | - | - |
| Definition: A finding based on lab | oratory test results that indicate in | creased levels of hemoglobin in a | biological specimen. | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>anticoagulation | >2.5 x ULN; >2.5 times above baseline if on anticoagulation | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the ratio of the patier | it's prothrombin time to a control s | ample in the blood. | |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of lipase in | a biological specimen. | | |
| _ymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of lymphocyte | es in a blood specimen. | | |
| _ymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormal increase in the numbe | r of lymphocytes in the blood, effu | sions or bone marrow. | |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of neutrophils | in a blood specimen. | | |
| Pancreatic enzymes decreased | <lln and="" asymptomatic<="" td=""><td>Increase in stool frequency,<br/>bulk, or odor; steatorrhea</td><td>Sequelae of absorption deficiency</td><td>-</td><td>-</td></lln> | Increase in stool frequency,<br>bulk, or odor; steatorrhea | Sequelae of absorption deficiency | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | 1 | ı<br>enzymes in a biological specimen. | • | • |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<="" 75,000="" <lln="" mm3;="" td=""><td>&lt;75,000 - 50,000/mm3; &lt;75.0 -</td><td>&lt;50,000 - 25,000/mm3; &lt;50.0 -</td><td>&lt;25,000/mm3; &lt;25.0 x 10e9 /L</td><td>-</td></lln> | <75,000 - 50,000/mm3; <75.0 - | <50,000 - 25,000/mm3; <50.0 - | <25,000/mm3; <25.0 x 10e9 /L | - |
| | 75.0 x 10e9 /L | 50.0 x 10e9 /L | 25.0 x 10e9 /L | | |
| Definition: A finding based on lab | poratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the levels of amylase | e in a serum specimen. | | |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | - |
| Definition: A finding based on tes | st results that indicate urine produc | ction is less relative to previous ou | tput. | • | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value; | <50% of predicted value; | - | - |
| | | limiting instrumental ADL | limiting self care ADL | | |
| Definition: A finding based on pu value. | lmonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | um inhalation) when compared to | the predicted |
| | 5 4400/ from honeling | 40 4000/ from honeling | >=20% from baseline | | |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | | - | 1- |
| | d by an increase in overall body w | 1 | · | 1 | |
| Weight loss | 5 to <10% from baseline; | 10 - <20% from baseline; | >=20% from baseline; tube | - | - |
| | intervention not indicated | nutritional support indicated | feeding or TPN indicated | | l |
| Definition: A finding characterize | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | T | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" td="" x<=""><td>&lt;3000 - 2000/mm3; &lt;3.0 - 2.0 x</td><td>&lt;2000 - 1000/mm3; &lt;2.0 - 1.0 x</td><td>&lt;1000/mm3; &lt;1.0 x 10e9 /L</td><td>-</td></lln> | <3000 - 2000/mm3; <3.0 - 2.0 x | <2000 - 1000/mm3; <2.0 - 1.0 x | <1000/mm3; <1.0 x 10e9 /L | - |
| | 10e9 /L | 10e9 /L | 10e9 /L | | |
| Definition: A finding based on lab | poratory test results that indicate a | n decrease in number of white blo | od cells in a blood specimen. | | |
| Investigations - Other, specify | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| cidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| efinition: A disorder characteriz | zed by abnormally high acidity (high | h hydrogen-ion concentration) of t | he blood and other body tissues. | | |
| Alcohol intolerance | - | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an increase in sensitivity to | the adverse effects of alcohol, wh | ich can include nasal congestion, | skin flushes, heart dysrhythmias, i | nausea, |
| romiting, indigestion and heada<br>Alkalosis | | | pH >7.5 | Life threatening consequences | Dooth |
| | pH >normal, but <=7.5 | <del>-</del><br> | 1. | Life-threatening consequences | Death |
| | zed by abnormally high alkalinity (lo | | | | l |
| Anorexia | Loss of appetite without alteration in eating habits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a loss of appetite. | | | | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | zed by excessive loss of water from | the body. It is usually caused by | severe diarrhea, vomiting or diaph | oresis. | |
| Glucose intolerance | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | zed by an inability to properly metal | bolize glucose. | | | |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | zed by laboratory test results that ir | ,<br>ndicate an elevation in the concen | ration of calcium (corrected for all | oumin) in blood. | • |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteriz<br>ntolerance. | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucose |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize the use of diuretic drugs. | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of potassium in the blood; a | associated with kidney failure or so | ometimes w |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23<br>mmol/L | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that in | ndicate an elevation in the concen | tration of magnesium in the blood | T | |
| lypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that in | | | T | T |
| lypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4 mmol/L;<br>life-threatening consequences | Death |
| efinition: A disorder characteriz | zed by laboratory test results that in | ndicate an elevation in the concen | | | 1 |
| lyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| efinition: A disorder characteriz | zed by laboratory test results that in | ndicate an elevation in the concen | tration of uric acid. | 1 | 1 |
| ypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by laboratory test results that ir | ndicate a low concentration of albu | ımin in the blood. | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -<br="">1.0 mmol/L</lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 - 6.0 mg/dL; <1.75 - 1.5 mmol/L; lonized calcium <0.9 - 0.8 mmol/L; hospitalization indicated | Corrected serum calcium of <6.0 mg/dL; <1.5 mmol/L; lonized calcium <0.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of calc | ium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0="" 55="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2<br/>mmol/L</td><td>&lt;40 - 30 mg/dL; &lt;2.2 - 1.7<br/>mmol/L</td><td>&lt;30 mg/dL; &lt;1.7 mmol/L; life-<br/>threatening consequences;<br/>seizures</td><td>Death</td></lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of gluc | ose in the blood. | · | _ |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><pre><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" pre="" symptomatic;=""></lln></pre></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <pre><lln -="" 3.0="" indicated<="" intervention="" l;="" mmol="" pre="" symptomatic;=""></lln></pre> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of pota | assium in the blood. | | |
| Hypomagnesemia | <lln -="" 0.5="" 1.2="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3<br/>mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3 mmol/L; life-<br/>threatening consequences</td><td>Death</td></lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of mag | gnesium in the blood. | | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of sod | ium in the blood. | | |
| Hypophosphatemia | <lln -="" 0.8="" 2.5="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL; &lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 - 1.0 mg/dL; &lt;0.6 - 0.3 mmol/L</td><td>&lt;1.0 mg/dL; &lt;0.3 mmol/L; life-<br/>threatening consequences</td><td>Death</td></lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6 mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3 mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of pho | sphates in the blood. | | |
| Iron overload | - | Moderate symptoms; intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by accumulation of iron in the t | issues. | | | |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| Definition: A disorder characteri | zed by having a high amount of boo | ly fat. | | | |
| Tumor lysis syndrome | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by metabolic abnormalities that | result from a spontaneous or the | rapy-related cytolysis of tumor cell | s. | |
| Metabolism and nutrition<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the abdomir | nal wall. | | |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in a joint. | 1 | Ī | |
| Arthritis | Mild pain with inflammation, erythema, or joint swelling | Moderate pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inflammation involving a joir | | 1 | | |
| Avascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by necrotic changes in the bon<br>ad the destruction of the bone struc | | od supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the back region. | | | |
| Bone pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the bones. | T | T | |
| Buttock pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the buttocks. | | | |
| Chest wall pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n in the chest wall region. | 1 | T | |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth | of bone. | | | |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characterize | ed by fibrotic degeneration of the | deep connective tissues. | 1 | , | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensatio | n on the lateral side of the body in | the region below the ribs and abo | ve the hip. | |
| Generalized muscle weakness | Symptomatic; weakness perceived by patient but not evident on physical exam | Symptomatic; weakness evident<br>on physical exam; weakness<br>limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | of muscles in multiple anatomic site | es. | T | |
| Growth suppression | Reduction in growth velocity by<br>10 - 29% ideally measured over<br>the period of a year | Reduction in growth velocity by 30 - 49% ideally measured over the period of a year or 0 - 49% reduction in growth from the baseline growth curve | Reduction in growth velocity of >=50% ideally measured over the period of a year | - | - |

| Musculoskeletal and connective tissue disorders Grade | | | | | |
|---|---|---|---|---|---|
| Advance Event | 1 | 2 | 3 | 4 | 5 |
| Adverse Event Head soft tissue necrosis | | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a necrotic process occurring | in the soft tissues of the head. | | | |
| Joint effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated; disabling | - | - |
| Definition: A disorder characterize | ed by excessive fluid in a joint, usu | ually as a result of joint inflammati | on. | T | 1 |
| Joint range of motion decreased | <=25% loss of ROM (range of motion); decreased ROM limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50% decrease in ROM; limiting self care ADL; disabling | - | - |
| Definition: A disorder characterize | ed by a decrease in joint flexibility | of any joint. | | | |
| Joint range of motion decreased cervical spine | Mild restriction of rotation or flexion between 60 - 70 degrees | Rotation <60 degrees to right or left; <60 degrees of flexion | Ankylosed/fused over multiple segments with no C-spine rotation | - | - |
| Definition: A disorder characterize | ed by a decrease in flexibility of a | cervical spine joint. | I | T | 1 |
| Joint range of motion decreased lumbar spine | Stiffness; difficulty bending to<br>the floor to pick up a very light<br>object but able to do athletic<br>activity | Pain with range of motion<br>(ROM) in lumbar spine; requires<br>a reaching aid to pick up a very<br>light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>ankylosis or fused over multiple<br>segments with no L-spine<br>flexion (e.g., unable to reach to<br>floor to pick up a very light<br>object) | - | - |
| Definition: A disorder characterize | ed by a decrease in flexibility of a | lumbar spine joint. | | | |
| Kyphosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an abnormal increase in the | curvature of the thoracic portion of | of the spine. | | |
| Lordosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an abnormal increase in the | curvature of the lumbar portion of | the spine. | | ı |
| Muscle weakness left-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characterize | ed by a reduction in the strength o | f the muscles on the left side of th | e body. | | |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characterize | ed by a reduction in the strength o | f the lower limb muscles. | | | |
| Muscle weakness right-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characterize | ed by a reduction in the strength o | f the muscles on the right side of t | the body. | ı | 1 |
| Muscle weakness trunk | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characterize | ed by a reduction in the strength o | f the trunk muscles. | | | |
| | | · | i | i | |

| Musculoskeletal and connective tissue disorders | | | | | |
|---|---|---|---|---|---|
| | Grade 1 2 3 4 5 | | | | |
| Adverse Event | 1 | 2 | | 4 | 5 |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g.,<br>shoe insert) or covered by<br>clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; disabling | - | - |
| Definition: A disorder characteri | zed by of a malformation of the mu | sculoskeletal system. | | | |
| Myalgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | | |
| Myositis | Mild pain | Moderate pain associated with weakness; pain limiting instrumental ADL | Pain associated with severe weakness; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by inflammation involving the s | keletal muscles. | | | |
| Neck pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the neck area. | T | | |
| Neck soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | g in the soft tissues of the neck. | | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of<br>osteoporosis or Bone Mineral<br>Density (BMD) t-score -1 to -2.5<br>(osteopenia); no loss of height<br>or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm;<br>hospitalization indicated; limiting<br>self care ADL | - | - |
| Definition: A disorder characteri composition), resulting in increa | zed by reduced bone mass, with a used fracture incidence. | decrease in cortical thickness and | in the number and size of the trab | peculae of cancellous bone (but no | ormal chemi |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the upper or lower extremities | ·<br>i. | | |
| Pelvic soft tissue necrosis | - zed by a necrotic process occurring | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Scoliosis | <20 degrees; clinically | | >45 dogrado: acapular | | |
| SCOIIOSIS | undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | | - |
| Definition: A disorder characteri | zed by a malformed, lateral curvatu | re of the spine. | 1 | <u> </u> | |
| Soft tissue necrosis lower limb | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | g in the soft tissues of the lower ex | tremity. | 1 | |
| Soft tissue necrosis upper limb | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |

| | Musculoskeletal and connective tissue disorders | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characterize | ed by fibrotic degeneration of the s | superficial soft tissues. | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, soft foods or purees | Decreased ROM with inability to adequately aliment or hydrate orally | - | - |
| Definition: A disorder characterize | ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | mastication. | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - 5 cm; shoe lift indicated; limiting instrumental ADL | , , | - | - |
| Definition: A disorder characterize | ed by of a discrepancy between th | e lengths of the lower or upper ex | tremities. | | |
| Musculoskeletal and connective tissue disorder - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Neoplasms benig | n, malignant and unspec | cified (incl cysts and poly | yps) | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Leukemia secondary to oncology chemotherapy | - | - | - | Present | Death |
| Definition: A disorder characterize | ed by leukemia arising as a result | of the mutagenic effect of chemot | herapy agents. | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by insufficiently healthy hemata | poietic cell production by the bone | e marrow. | | |
| Treatment related secondary malignancy | - | - | Non life-threatening secondary malignancy | Acute life-threatening secondary malignancy; blast crisis in leukemia | Death |
| Definition: A disorder characterize | ed by development of a malignand | by most probably as a result of trea | atment for a previously existing ma | alignancy. | |
| Tumor pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort from a ne | eoplasm that may be pressing on | a nerve, blocking blood vessels, ir | nflamed or fractured from metastas | sis. |
| Neoplasms benign, malignant<br>and unspecified (incl cysts and<br>polyps) - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Nervous system disorders | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abducens nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by involvement of the abducen | s nerve (sixth cranial nerve). | 1 | I | 1 |
| Accessory nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the accessor | ry nerve (eleventh cranial nerve). | | <b>-</b> | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the acoustic | nerve (eighth cranial nerve). | | T | |
| Akathisia | Mild restlessness or increased motor activity | Moderate restlessness or increased motor activity; limiting instrumental ADL | Severe restlessness or increased motor activity; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by an uncomfortable feeling of | inner restlessness and inability to | stay still; this is a side effect of so | me psychotropic drugs. | |
| Amnesia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss;<br>limiting self care ADL | - | - |
| | zed by systematic and extensive lo | ss or memory. | V-: | | T |
| Aphonia | - | - | Voicelessness; unable to speak | 1 | 1- |
| Definition: A disorder characteriz | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by inflammation of the arachno | id membrane and adjacent subara | achnoid space. | | |
| Ataxia | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | - | - |
| Definition: A disorder characteriz | zed by lack of coordination of musc | ।<br>ale movements resulting in the imp | 1 | ı<br>ıntarv activities. | 1 |
| Brachial plexopathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by regional paresthesia of the l | brachial plexus, marked discomfor | t and muscle weakness, and limite | ed movement in the arm or hand. | |
| Central nervous system<br>necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms;<br>corticosteroids indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a necrotic process occurring | in the brain and/or spinal cord. | 1 | I | , |
| Cerebrospinal fluid leakage | Post-craniotomy: asymptomatic;<br>Post-lumbar puncture: transient<br>headache; postural care<br>indicated | Post-craniotomy: moderate<br>symptoms; medical intervention<br>indicated; Post-lumbar<br>puncture: persistent moderate<br>symptoms; blood patch<br>indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by loss of cerebrospinal fluid in | to the surrounding tissues. | T | T | |
| Cognitive disturbance | Mild cognitive disability; not<br>interfering with work/school/life<br>performance; specialized<br>educational services/devices<br>not indicated | Moderate cognitive disability;<br>interfering with work/school/life<br>performance but capable of<br>independent living; specialized<br>resources on part time basis<br>indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | - | - |
| Definition: A disorder characterize | zed by a conspicuous change in co | gnitive function. | 1 | T | |
| Concentration impairment | Mild inattention or decreased level of concentration | Moderate impairment in attention or decreased level of concentration; limiting instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | - | - |

| Nervous system disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to stimuli; limiting instrumental ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by a decrease in ability to perc | eive and respond. | | | 1 |
| Dizziness | Mild unsteadiness or sensation of movement | Moderate unsteadiness or sensation of movement; limiting instrumental ADL | Severe unsteadiness or sensation of movement; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a disturbing sensation of ligi | htheadedness, unsteadiness, gidd | iness, spinning or rocking. | | |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characteriz | ed by slow and slurred speech res | sulting from an inability to coordina | te the muscles used in speech. | T | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation. | T | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet<br>(e.g., oral supplements);<br>noxious or unpleasant taste;<br>loss of taste | - | - | - |
| Definition: A disorder characteriz | ed by abnormal sensual experienc | ce with the taste of foodstuffs; it ca | n be related to a decrease in the | sense of smell. | |
| Dysphasia | Awareness of receptive or expressive characteristics; not impairing ability to communicate | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | - | - |
| Definition: A disorder characteriz | ed by impairment of verbal commu | unication skills, often resulting fron | n brain damage. | 1 | |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | - |
| Definition: A disorder characteriz | ed by swelling due to an excessive | e accumulation of fluid in the brain | T | T | |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a pathologic process involvi | ng the brain. | <u> </u> | <u> </u> | 1 |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary movements; limiting instrumental ADL | Severe involuntary movements or torticollis; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by abnormal, repetitive, involur | ntary muscle movements, frenzied | speech and extreme restlessness | <b>5.</b> | |
| Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | of the facial muscles. | <u> </u> | <u> </u> | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the facial ne | rve (seventh cranial nerve). | | | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the glossoph | aryngeal nerve (ninth cranial nerv | e). | | |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in various parts of the head | not confined to the area of distrib | ution of any nerve. | 1 |
| Hydrocephalus | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; intervention not indicated | Severe symptoms or neurological deficit; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal increase of cer | rebrospinal fluid in the ventricles o | f the brain. | 1 | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | - | - |

| Nervous system disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypoglossal nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | | | |
| Definition: A disorder characteriz | zed by involvement of the hypoglos | sal nerve (twelfth cranial nerve). | T | T | |
| Intracranial hemorrhage | Asymptomatic; clinical or | Moderate symptoms; medical | Ventriculostomy, ICP | Life-threatening consequences; | Death |
| | diagnostic observations only; | intervention indicated | monitoring, intraventricular | urgent intervention indicated | |
| | intervention not indicated | | thrombolysis, or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characterize | zed by bleeding from the cranium. | I | T | T | |
| Ischemia cerebrovascular | Asymptomatic; clinical or | Moderate symptoms | - | - | - |
| | diagnostic observations only; | | | | |
| | intervention not indicated | | | | |
| Definition: A disorder characteriz | zed by a decrease or absence of bl | ood supply to the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | ological |
| damage. | | | | | |
| IVth nerve disorder | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | diagnostic observations only; | instrumental ADL | care ADL | | |
| | intervention not indicated | | | | |
| Definition: A disorder characterize | zed by involvement of the trochlear | nerve (fourth cranial nerve). | • | • | • |
| | Mild symptoms; reduced | Moderate symptoms; limiting | _ | _ | |
| Lethargy | alertness and awareness | instrumental ADL | | | - |
| Definition: A disease to the control of the control | 1 | 1 | <br> | I | I |
| Definition: A disorder characterize | zed by a decrease in consciousnes | s characterized by mental and phy | ysical inertness.<br>I | 1 | |
| Leukoencephalopathy | Asymptomatic; small focal | Moderate symptoms; focal | Severe symptoms; extensive | Life-threatening consequences; | Death |
| | T2/FLAIR hyperintensities; | T2/FLAIR hyperintensities, | T2/FLAIR hyperintensities, | extensive T2/FLAIR | |
| | involving periventricular white | involving periventricular white | involving periventricular white | hyperintensities, involving | |
| | matter or <1/3 of susceptible | matter extending into centrum | matter involving 2/3 or more of | periventricular white matter | |
| | areas of cerebrum +/- mild | semiovale or involving 1/3 to 2/3 | susceptible areas of cerebrum | involving most of susceptible | |
| | increase in subarachnoid space | of susceptible areas of | +/- moderate to severe increase | areas of cerebrum +/- moderate | |
| | (SAS) and/or mild | cerebrum +/- moderate increase | in SAS and/or moderate to | to severe increase in SAS | |
| | ventriculomegaly | in SAS and/or moderate | severe ventriculomegaly | and/or moderate to severe | |
| | | ventriculomegaly | | ventriculomegaly | |
| Definition: A disorder characteriz | zed by diffuse reactive astrocytosis | with multiple areas of necrotic foo | ci without inflammation. | | |
| Memory impairment | Mild memory impairment | Moderate memory impairment; | Severe memory impairment; | - | _ |
| , , | , , | limiting instrumental ADL | limiting self care ADL | | |
| Definition: A disorder characteriz | red by a deterioration in memory fu | - | | 1 | |
| | | | C | Life the extension | D 41- |
| Meningismus | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | I | instrumental ADL | care ADL | urgent intervention indicated | l |
| Definition: A disorder characterize | zed by neck stiffness, headache, a | nd photophobia resulting from irrita | ation of the cerebral meninges. | 1 | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| | | instrumental ADL | care ADL | | |
| Definition: A disorder characteriz | zed by uncontrolled and purposeles | ss movements. | | | |
| Myelitis | Asymptomatic; mild signs (e.g., | Moderate weakness or sensory | Severe weakness or sensory | Life-threatening consequences; | Death |
| , 511110 | Babinski's reflex or Lhermitte's | loss; limiting instrumental ADL | loss; limiting self care ADL | urgent intervention indicated | Boaut |
| | sign) | | | a. gont into vondon indicated | |
| Definition: A disorder sharest | 1 | ninal cord. Symptoms in aluda ···- | kness parasthosia semesul | marked discomfort and incention | l<br>nce |
| | zed by inflammation involving the s | | T . | marked discomion and incontiner | ice. |
| Neuralgia | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characterize | zed by intense painful sensation alo | ong a nerve or group of nerves. | 1 | 1 | |
| Nystagmus | - | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| - | | instrumental ADL | care ADL | | |
| Definition: A disorder characterize | zed by involuntary movements of th | ne eyeballs. | | • | • |
| Oculomotor nerve disorder | | | Covere symptoms: limiting If | | |
| | Asymptomatic; clinical or | Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |
| Oculoritotol Herve disorder | diagnostic observations only; | instrumental ADL | care ADL | | |
| Occioniotol herve disorder | | İ | 1 | 1 | 1 |
| | intervention not indicated | | | | |
| | Intervention not indicated zed by involvement of the oculomo | tor nerve (third cranial nerve). | 1 | 1 | |
| | 1 | or nerve (third cranial nerve). Moderate symptoms; limiting | Severe symptoms; limiting self | - | - |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize are experienced in the absence of | | ensory neurons resulting in abnorr | mal cutaneous sensations of tinglin | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation or degeneration | on of the peripheral motor nerves. | | | |
| Peripheral sensory neuropathy | Asymptomatic; loss of deep tendon reflexes or paresthesia | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation or degeneratio | on of the peripheral sensory nerves | S. | | |
| Phantom pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort related to | o a limb or an organ that is remove | ed from or is not physically part of | the body. | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| Definition: A disorder characterize | ed by an episode of lightheadedne | ess and dizziness which may prec | ede an episode of syncope. | T | |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by dysfunction of the corticospi<br>nd a decrease in fine motor coord | | I cord. Symptoms include an incre | ease in the muscle tone in the lower | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting instrumental ADL; medical intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize connecting nerve root. | ed by inflammation involving a ner | rve root. Patients experience mark | led discomfort radiating along a ne | rve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by paralysis of the recurrent lar | ryngeal nerve. | | | |
| Reversible posterior<br>leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very<br>abnormal imaging studies;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | - | = | | indings of posterior leukoencephal<br>s an acute or subacute reversible o | |
| Seizure | Brief partial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characterize | ed by a sudden, involuntary skelet | tal muscular contractions of cerebi | ral or brain stem origin. | | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort in the fac | ce, between the eyes, or upper tee | eth originating from the sinuses. | | |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by characterized by excessive | sleepiness and drowsiness. | | | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle tone and increase in resistance through range of motion | Severe increase in muscle tone and increase in resistance through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characterized disturbances. | ed by increased involuntary muscl | | | It results in gait, movement, and sp | peech |
| Stroke | Asymptomatic or mild neurologic deficit; radiographic findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a sudden loss of sensory fu | nction due to an intracranial vascu | ılar event. | 1 | |
| Syncope | - | - | Fainting; orthostatic collapse | - | - |
| Definition: A disorder characterize | ed by spontaneous loss of consci | ousness caused by insufficient blo | od supply to the brain. | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with or without imaging confirmation | - | - | - |
| Definition: A disorder characteriz | ed by a brief attack (less than 24 h | nours) of cerebral dysfunction of va | ascular origin, with no persistent n | eurological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by the uncontrolled shaking mo | vement of the whole body or indiv | ridual parts. | | |
| Trigeminal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by involvement of the trigemina | l nerve (fifth cranial nerve). | | | |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by involvement of the vagus ne | rve (tenth cranial nerve). | • | | |
| Vasovagal reaction | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz increase in the stimulation of the | ed by a sudden drop of the blood progressing vagus nerve. | oressure, bradycardia, and periph | eral vasodilation that may lead to | loss of consciousness. It results fr | om an |
| Nervous system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Pregna | ancy, puerperium and pe | rinatal conditions | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Fetal death | - | - | - | - | Fetal loss at<br>any<br>gestational<br>age |
| Definition: A disorder characterize | ed by death in utero; failure of the | product of conception to show evi | idence of respiration, heartbeat, or | definite movement of a voluntary | muscle after |
| expulsion from the uterus, withou | t possibility of resuscitation. | | | | |
| Fetal growth retardation | - | <10% percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | - |
| Definition: A disorder characterize | ed by inhibition of fetal growth resu | ulting in the inability of the fetus to | achieve its potential weight. | | |
| Premature delivery | Delivery of a liveborn infant at >34 to 37 weeks gestation | Delivery of a liveborn infant at >28 to 34 weeks gestation | Delivery of a liveborn infant at 24 to 28 weeks gestation | Delivery of a liveborn infant at 24 weeks of gestation or less | - |
| Definition: A disorder characterize gestation. | ed by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | tween the twentieth and thirty-sev | enth week of |
| Unintended pregnancy | - | - | Unintended pregnancy | - | - |
| Definition: A disorder characterize | ed by an unexpected pregnancy a | t the time of conception. | | | · |
| Pregnancy, puerperium and perinatal conditions - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing | Life-threatening consequences; urgent intervention indicated | Death |
| | | | hospitalization indicated;<br>disabling; limiting self care ADL | | |

| | | Psychiatric disor | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation; hospitalization not indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by a state of restlessness asso | | irritability and tension. | | |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| | erized by an inability to achieve orgas | | | | |
| Anxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization not indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder characte stimulus. | erized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dys | pnea unattached to a clearly iden | tifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by a lack of clear and orderly the | nought and behavior. | | | |
| Delayed orgasm | | Delay in achieving orgasm adversely affecting relationship | - | - | - |
| | erized by sexual dysfunction characte | | T | I | I_ |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder character reversible condition. | erized by the acute and sudden devel | opment of confusion, illusions, mo | ovement changes, inattentiveness, | agitation, and hallucinations. Usu | ally, it is a |
| Delusions | - | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by false personal beliefs held c | ontrary to reality, despite contradi | ctory evidence and common sense | e. | |
| Depression | Mild depressive symptoms | Moderate depressive symptoms; limiting instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by melancholic feelings of grief | or unhappiness. | ' | ' | • |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | - |
| Definition: A disorder characte | erized by an exaggerated feeling of w | ell-being which is disproportionate | to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | Death |
| Definition: A disorder characte | erized by a false sensory perception i | n the absence of an external stimu | ılus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling asleep, staying asleep or waking up early | - | - |
| Definition: A disorder characte | erized by difficulty in falling asleep an | d/or remaining asleep. | | | |
| Libido decreased | Decrease in sexual interest not adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by a decrease in sexual desire | T | 1 | T | 1 |
| Libido increased | Mild increase in sexual interest not adversely affecting relationship | Moderate increase in sexual interest adversely affecting relationship | Severe increase in sexual interest leading to dangerous behavior | - | - |
| Definition: A disorder characte | erized by an increase in sexual desire | ). | | | |
| Mania | Mild manic symptoms (e.g.,<br>elevated mood, rapid thoughts,<br>rapid speech, decreased need<br>for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by excitement of psychotic prop | oortions manifested by mental and | l physical hyperactivity, disorganiz | ation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |

| | | Psychiatric disord | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | ed by a conspicuous change in a p | person's behavior and thinking. | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characteriz tumor. | ed by personality change, impaire | d functioning, and loss of touch wi | th reality. It may be a manifestatio | n of schizophrenia, bipolar disorde | er or brain |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an inability to rest, relax or b | pe still. | | | |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide<br>with serious intent to die which<br>requires hospitalization | - |
| Definition: A disorder characteriz | ed by thoughts of taking one's owr | n life. | | | |
| Suicide attempt | - | - | Suicide attempt or gesture without intent to die which may not require hospitalization | Suicide attempt with intent to die which requires hospitalization | Death |
| Definition: A disorder characteriz | ed by self-inflicted harm in an atte | mpt to end one's own life. | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |

| Renal and urinary disorders | | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute kidney injury Definition: A disorder character | Creatinine level increase of >0.3 mg/dL; creatinine 1.5 - 2.0 x above baseline ized by the acute loss of renal functions. | baseline | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated | Life-threatening consequences;<br>dialysis indicated | Death |
| causes (ureteral or bladder out | • | , | | ,,, | |
| Bladder perforation | - | Extraperitoneal perforation, indwelling catheter indicated | Intraperitoneal perforation;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>organ failure; urgent operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by a rupture in the bladder wall | | 1 | <u> </u> | |
| Bladder spasm | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | - | - |
| Definition: A disorder character | ized by a sudden and involuntary co | ontraction of the bladder wall. | | | |
| Chronic kidney disease | eGFR (estimated Glomerular<br>Filtration Rate) or CrCl<br>(creatinine clearance) <lln -="" 60<br="">ml/min/1.73 m2 or proteinuria<br/>2+ present; urine<br/>protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15 ml/min/1.73 m2; dialysis or renal transplant indicated | Death |
| Definition: A disorder character | ized by gradual and usually perman | ent loss of kidney function resulting | ng in renal failure. | <b>-</b> | |
| Cystitis noninfective | Microscopic hematuria; minimal increase in frequency, urgency, dysuria, or nocturia; new onset of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV<br>medications or hospitalization<br>indicated; elective endoscopic,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the bladder | ,<br>which is not caused by an infectio | n of the urinary tract. | • | |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate blood in the urine. | | | |
| Hemoglobinuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate the presence of free hemo | globin in the urine. | | |
| Proteinuria | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 - 3.4 g/24 hrs;<br>Pediatric: urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5<br>g/24 hrs;<br>Pediatric: urine P/C >1.9 | - | - |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate the presence of excessive | protein in the urine. It is predomin | antly albumin, but also globulin. | |
| Renal calculi | Asymptomatic or mild symptoms; occasional use of nonprescription analgesics indicated | Symptomatic; oral antiemetics indicated; around the clock nonprescription analgesics or any oral narcotic analgesics indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences;<br>urgent radiologic, endoscopic or<br>operative intervention indicated | Death |
| Definition: A disorder character | ized by the formation of crystals in t | he pelvis of the kidney. | | | |
| Renal colic | Mild pain not interfering with activity; nonprescription medication indicated | Moderate pain; limiting instrumental ADL; prescription medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |

| | | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or hospitalization indicated; elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the kidney. | | | | |
| Urinary fistula | - | Noninvasive intervention indicated; urinary or suprapubic catheter placement indicated | Limiting self care ADL; elective<br>radiologic, endoscopic or<br>operative intervention indicated;<br>permanent urinary diversion<br>indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between any part of the urinary s | system and another organ or anato | omic site. | |
| Urinary frequency | Present | Limiting instrumental ADL;<br>medical management indicated | - | - | - |
| Definition: A disorder characteriz | ed by urination at short intervals. | | _ | | |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inability to control the flow o | f urine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by accumulation of urine within | the bladder because of the inabil | ity to urinate. | | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ<br>function (e.g., hydronephrosis,<br>or renal dysfunction); elective<br>radiologic, endoscopic or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of contents of the urinary tract. | | | |
| Urinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the urinary tract. | | | |
| Urinary urgency | Present | Limiting instrumental ADL; medical management indicated | - | - | - |
| Definition: A disorder characteriz | ed by a sudden compelling urge to | urinate. | | | |
| Urine discoloration | Present | - | - | - | - |
| Definition: A disorder characteriz | ed by a change in the color of the | urine. | | | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azoospermia | - | - | Absence of sperm in ejaculate | - | - |
| Definition: A disorder characte | erized by laboratory test results that in | ndicate complete absence of speri | natozoa in the semen. | | |
| Breast atrophy | Minimal asymmetry; minimal | Moderate asymmetry; moderate | Asymmetry >1/3 of breast | - | - |
| . , | atrophy | atrophy | volume; severe atrophy | | |
| Definition: A disorder characte | erized by underdevelopment of the br | east. | | | , |
| Breast pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| • | | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by marked discomfort sensation | n in the breast region. | | | ` |
| Dysmenorrhea | Mild symptoms; intervention not | Moderate symptoms; limiting | Severe symptoms; limiting self | - | _ |
| , | indicated | instrumental ADL | care ADL | | |
| Definition: A disorder characte | rized by abnormally painful abdomin | al cramps during menses. | ! | ' | • |
| Dyspareunia | Mild discomfort or pain | Moderate discomfort or pain | Severe discomfort or pain | _ | _ |
| 3 yopar ourna | associated with vaginal | associated with vaginal | associated with vaginal | | |
| | penetration; discomfort relieved | penetration; discomfort or pain | penetration; discomfort or pain | | |
| | with use of vaginal lubricants or | partially relieved with use of | unrelieved by vaginal lubricants | | |
| | estrogen | vaginal lubricants or estrogen | or estrogen | | |
| Definition: A disorder characte | rized by painful or difficult coitus. | | | | |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde | - | - | - |
| | | ejaculation | | | |
| Definition: A disorder characte | rized by problems related to ejaculat | ion. This category includes prema | ture, delayed, retrograde and pair | ful ejaculation. | |
| Erectile dysfunction | Decrease in erectile function | Decrease in erectile function | Decrease in erectile function | - | _ |
| , | (frequency or rigidity of | (frequency/rigidity of erections), | (frequency/rigidity of erections) | | |
| | erections) but intervention not | erectile intervention indicated, | but erectile intervention not | | |
| | indicated (e.g., medication or | (e.g., medication or mechanical | helpful (e.g., medication or | | |
| | use of mechanical device, | devices such as penile pump) | mechanical devices such as | | |
| | penile pump) | | penile pump); placement of a | | |
| | | | permanent penile prosthesis | | |
| | | | indicated (not previously present) | | |
| D-6:iti | | | | l | 1 |
| | erized by the persistent or recurrent in | | | | T |
| Fallopian tube obstruction | Diagnostic observations only; | Mild symptoms; elective | Severe symptoms; elective | - | - |
| | intervention not indicated | intervention indicated | operative intervention indicated | | l |
| Definition: A disorder characte | erized by blockage of the normal flow | of the contents in the fallopian tub | oe.<br>T | | |
| Fallopian tube stenosis | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| | diagnostic observations only; | not indicated | operative intervention indicated | urgent operative intervention | |
| | intervention not indicated | | | indicated (e.g., organ resection) | |
| Definition: A disorder characte | erized by a narrowing of the fallopian | tube lumen. | T | I | 1 |
| Female genital tract fistula | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| | diagnostic observations only; | not indicated | operative intervention indicated | urgent intervention indicated | |
| | intervention not indicated | | | | |
| Definition: A disorder characte | rized by an abnormal communication | between a female reproductive s | ystem organ and another organ o | r anatomic site. | _ |
| Feminization acquired | Mild symptoms; intervention not | Moderate symptoms; medical | - | - | - |
| | indicated | intervention indicated | | | |
| Definition: A disorder characte | erized by the development of secondar | ary female sex characteristics in m | ales due to extrinsic factors. | | |
| Genital edema | Mild swelling or obscuration of | Readily apparent obscuration of | Lymphorrhea; gross deviation | - | - |
| | anatomic architecture on close | anatomic architecture; | from normal anatomic contour; | | |
| | inspection | obliteration of skin folds; readily | limiting self care ADL | | |
| | | apparent deviation from normal | | | |
| | | anatomic contour | l | | I |
| Definition: A disorder characte | erized by swelling due to an excessive | e accumulation of fluid in the genit | als. | 1 | |
| Gynecomastia | Asymptomatic breast | Symptomatic (e.g., pain or | Severe symptoms; elective | - | - |
| | enlargement | psychosocial impact) | operative intervention indicated | | |
| Definition: A disorder characte | erized by excessive development of the | ne breasts in males. | | | |
| -lematosalpinx | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| •<br>• | imaging study or laparoscopy; | intervention indicated | indicated; radiologic or | urgent operative intervention | |
| | intervention not indicated | | endoscopic intervention | indicated | |
| | Rep | productive system and bi | reast disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteri | zed by the presence of blood in a fa | allopian tube. | | | |
| rregular menstruation | Intermittent menses with skipped menses for no more than 1 to 3 months | Intermittent menses with skipped menses for more than 4 to 6 months | Persistent amenorrhea for more than 6 months | - | - |
| Definition: A disorder characteri | zed by irregular cycle or duration of | f menses. | I | I | |
| actation disorder | Mild changes in lactation, not<br>significantly affecting production<br>or expression of breast milk | Changes in lactation,<br>significantly affecting breast<br>production or expression of<br>breast milk | - | - | - |
| Definition: A disorder characteri | zed by disturbances of milk secretion | on. It is not necessarily related to p | pregnancy that is observed in fema | ales and can be observed in males | S. |
| Menorrhagia | Mild; iron supplements indicated | Moderate symptoms; medical intervention indicated (e.g., hormones) | Severe; transfusion indicated;<br>surgical intervention indicated<br>(e.g., hysterectomy) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by abnormally heavy vaginal bl | eeding during menses. | | | |
| Nipple deformity | Asymptomatic; asymmetry with slight retraction and/or thickening of the nipple areolar complex | Symptomatic; asymmetry of<br>nipple areolar complex with<br>moderate retraction and/or<br>thickening of the nipple areolar<br>complex | - | - | - |
| Definition: A disorder characteri | zed by a malformation of the nipple | | | | |
| Oligospermia | Sperm concentration >48 million/mL or motility >68% | Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Sperm concentration <13 million/mL or motility <32% | - | - |
| Definition: A disorder characteri | zed by a decrease in the number of | spermatozoa in the semen. | | | |
| Ovarian hemorrhage | Minimal bleeding identified on<br>imaging study or laproscopy;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the ovary. | • | ' | ' | • |
| Ovarian rupture | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by tearing or disruption of the c | varian tissue. | , . | | ' |
| Ovulation pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri<br>ovarian follicle. | zed by marked discomfort sensatio | n in one side of the abdomen betw | veen menstrual cycles, around the | time of the discharge of the ovum | from the |
| Pelvic floor muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic, not interfering<br>with bladder, bowel, or vaginal<br>function; limiting instrumental<br>ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a reduction in the strength o | f the muscles of the pelvic floor. | | | _ |
| elvic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the pelvis. | T | I | T |
| Penile pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | zed by marked discomfort sensatio | | I | | |
| erineal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the area between the ger | 1 | Т | |
| Premature menopause | - | - | Present | - | - |
| Definition: A disorder characteri | zed by ovarian failure before the ag | je of 40. Symptoms include hot fla | shes, night sweats, mood swings | and a decrease in sex drive. | |
| Prostatic hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Rep | productive system and be | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | zed by bleeding from the prostate of | land. | 1 | | |
| Prostatic obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz<br>tream, and incomplete emptyin | zed by compression of the urethra g of the bladder). | secondary to enlargement of the p | prostate gland. This results in voidi | ng difficulties (straining to void, sl | ow urine |
| Prostatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | omfort in the prostate gland. | | | |
| Scrotal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by marked discomfort sensatio | n in the scrotal area. | | | |
| Spermatic cord hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the spermatic | cord. | | | |
| Spermatic cord obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the contents of the spermatic c | ord. | | |
| Festicular disorder | Asymptomatic; clinical or diagnostic observations only; | Symptomatic but not interfering with urination or sexual | Severe symptoms; interfering with urination or sexual function; | Life-threatening consequences; urgent intervention indicated | Death |
| | intervention not indicated | activities; intervention not indicated; limiting instrumental ADL | limiting self care ADL;<br>intervention indicated | | |
| Definition: A disorder characteriz | zed by involvement of the testis. | I | 1 | I | ı |
| Testicular hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the testis. | 1 | 1 | | |
| esticular pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | zed by a sensation of marked disco | omfort in the testis. | | T | |
| Jterine fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | red by an abnormal communication | n between the uterus and another | organ or anatomic site. | I | 1 |
| Jterine hemorrhage | | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by bleeding from the uterus. | ' | | • | |
| Iterine obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | zed by blockage of the uterine outle | et. | | | |
| Iterine pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| efinition: A disorder characteriz | zed by a sensation of marked disco | omfort in the uterus. | 1 | | |
| /aginal discharge | Mild vaginal discharge (greater than baseline for patient) | Moderate to heavy vaginal discharge; use of perineal pad or tampon indicated | - | - | - |
| Definition: A disorder characterize | ा<br>zed by vaginal secretions. Mucus p | | discharged from the vagina natura | lly, especially during the childbea | ring years. |
| /aginal dryness | Mild vaginal dryness not interfering with sexual function | Moderate vaginal dryness interfering with sexual function | Severe vaginal dryness resulting in dyspareunia or severe discomfort | - | - |
| Definition: A disorder characteriz | l<br>zed by an uncomfortable feeling of | or causing frequent discomfort itching and burning in the vagina. | 1557010 dissolition | I<br> | I |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between the vagina and another | organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on<br>clinical exam or imaging study;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema, or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal ulceration; life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation involving the v | agina. Symptoms may include red | lness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characterize | ed by blockage of vaginal canal. | | 1 | 1 | |
| Vaginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | mfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ·<br>ed by a rupture in the vaginal wall. | | • | • | • |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or<br>shortening not interfering with<br>physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characterize | ed by a narrowing of the vaginal c | anal. | | | _ |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | - | - |
| Definition: A disorder characterize intercourse. | ed by involuntary spasms of the po | elvic floor muscles, resulting in pa | thologic tightness of the vaginal w | all during penetration such as duri | ng sexual |
| Reproductive system and breast disorders - Other, specify | * ' | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | I | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adult respiratory distress<br>syndrome | - | - | Present with radiologic findings; intubation not indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri<br>surgery. | zed by progressive and life-threater | ning pulmonary distress in the abs | ence of an underlying pulmonary | condition, usually following major t | rauma or |
| Allergic rhinitis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| | zed by an inflammation of the nasa<br>s of the sinuses, eyes, middle ear, a | • | • | • | ay also |
| Apnea | - | - | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by cessation of breathing. | T | I | T | |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Altered eating habits; coughing or choking episodes after eating or swallowing; medical intervention indicated (e.g., suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or hemodynamic compromise; intubation or urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by inhalation of solids or liquids | s into the lungs. | | <u> </u> | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by the collapse of part or the en | ntire lung. | T | T | 1 |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube thoracostomy or medical management indicated; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | · | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild<br>wheezing); endoscopic<br>evaluation indicated;<br>radiographic evidence of<br>atelectasis/lobar collapse;<br>medical management indicated<br>(e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by blockage of a bronchus pas | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor;<br>endoscopic intervention<br>indicated (e.g., laser, stent<br>placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | zed by a narrowing of the bronchial | 1 | | leg at the second | <b>.</b> |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between a bronchus and the ple | ural cavity. | I | |
| Bronchopulmonary hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g., | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention | Death |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bronchospasm | Mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Limiting self care ADL; oxygen saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a sudden contraction of the | smooth muscles of the bronchial | wall. | 1 | 1 |
| Chylothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thoracentesis or tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | rized by milky pleural effusion (abnor | rmal collection of fluid) resulting fr | om accumulation of lymph fluid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription intervention indicated | Moderate symptoms, medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte by a distinctive sound. | rized by sudden, often repetitive, spa | asmodic contraction of the thoraci | c cavity, resulting in violent release | e of air from the lungs and usually | accompanie |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an uncomfortable sensation | of difficulty breathing. | | | |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; topical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the nose. | l | T | 1 | |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe symptoms; interfering with sleep; limiting self care ADL | - | - |
| | rized by repeated gulp sounds that re | | | ttributed to a spasm of the diaphra | igm. |
| Hoarseness | Mild or intermittent voice change; fully understandable; self-resolves | Moderate or persistent voice changes; may require occasional repetition but understandable on telephone; medical evaluation indicated | Severe voice changes including predominantly whispered speech | - | - |
| Definition: A disorder characte | rized by harsh and raspy voice arisin | g from or spreading to the larynx. | | | |
| Нурохіа | - | Decreased oxygen saturation<br>with exercise (e.g., pulse<br>oximeter <88%); intermittent<br>supplemental oxygen | Decreased oxygen saturation at rest (e.g., pulse oximeter <88% or PaO2 <=55 mm Hg) | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characte | rized by a decrease in the level of ox | tygen in the body. | 1 | 1 | 1 |
| Laryngeal edema | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | Stridor; respiratory distress;<br>hospitalization indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | rized by swelling due to an excessive | , | | Life ii. | D 11 |
| Laryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the larynx and another | organ or anatomic site. | | |
| Laryngeal hemorrhage | Mild cough or trace hemoptysis; laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characte | rized by bleeding from the larynx. | ī | T | ī | ı |

| | | ratory, thoracic and med | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| aryngeal mucositis | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered oral intake | Severe pain; severely altered eating/swallowing; medical intervention indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characteriz | ed by an inflammation involving th | e mucous membrane of the larynx | ·<br>(. | • | • |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the laryngeal ai | way. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a narrowing of the laryngeal | | Causes as mentames disappea and | Life threatening concessions | Dooth |
| Laryngopharyngeal dysesthesia | Mild symptoms; no anxiety; intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and swallowing difficulty; limiting self care ADL | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by an uncomfortable persistent | sensation in the area of the laryn | gopharynx. | | |
| Laryngospasm | - | Transient episode; intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characteriz | ।<br>ed by paroxysmal spasmodic mus | I<br>cular contraction of the vocal cord | | Interpretation Detect in Jeouetry | l |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical | Transfusion, radiologic, endoscopic, or elective operative intervention indicated (e.g., hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the mediastin | um. | | <b>,</b> | |
| Nasal congestion | Mild symptoms; intervention not indicated | intervention indicated | Associated with bloody nasal discharge or epistaxis | - | - |
| | ed by obstruction of the nasal pas | | | | l |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the pharynx and anothe | er organ or anatomic site. | <del> </del> | |
| Pharyngeal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the pharynx. | Moderate pain and analysis: | Sovere pain: unable to | Life threatening assessment | Death |
| Pharyngeal mucosius | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics indicated; altered oral intake; limiting instrumental ADL | Severe pain; unable to adequately aliment or hydrate orally; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an inflammation involving th | e mucous membrane of the phary | rnx. | Γ | ı |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Respir | ratory, thoracic and med | lastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | rized by a necrotic process occurring | in the pharynx. | 1 | 1 | |
| Pharyngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder character | rized by a narrowing of the pharynge | al airway. | ' | ' | ' |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by marked discomfort sensation | n in the pharyngolaryngeal region. | | <u> </u> | ı |
| Pleural effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., diuretics or limited therapeutic thoracentesis) | Symptomatic with respiratory<br>distress and hypoxia; surgical<br>intervention including chest tube<br>or pleurodesis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | rized by an increase in amounts of flo | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or associated with pneumothorax; chest tube drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | rized by bleeding from the pleural ca | vity. | • | • | • |
| Pleuritic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by marked discomfort sensation | n in the pleura. | T | T | |
| Pneumonitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | rized by inflammation focally or diffus | | | | I |
| Pneumothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative intervention indicated; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by abnormal presence of air in | the pleural cavity resulting in the | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | rized by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | |
| Productive cough | | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | - | - |
| | rized by expectorated secretions upo | | Covere diannes er diannes et | Life threatening requireten. | Dooth |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at rest; oxygen indicated; limiting self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder character | rized by accumulation of fluid in the I | | nce of the gas exchange that may | lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia; radiologic<br>pulmonary fibrosis <25% of lung<br>volume | Moderate hypoxemia; evidence<br>of pulmonary hypertension;<br>radiographic pulmonary fibrosis<br>25 - 50% | Severe hypoxemia; evidence of right-sided heart failure; radiographic pulmonary fibrosis >50 - 75% | Life-threatening consequences (e.g., hemodynamic/pulmonary complications); intubation with ventilatory support indicated; radiographic pulmonary fibrosis >75% with severe honeycombing | Death |
| Definition: A disorder character | rized by the replacement of the lung | tissue by connective tissue, leadir | ng to progressive dyspnea, respira | tory failure or right heart failure. | |
| Pulmonary fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| | Respi | ratory, thoracic and med | astinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | red by an abnormal communication | between the lung and another or | gan or anatomic site. | <u> </u> | |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other evaluation | Moderate dyspnea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated<br>with hypoxemia, right heart<br>failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | ed by an increase in pressure with | in the pulmonary circulation due to | lung or heart disorder. | | |
| Respiratory failure | - | - | - | Life-threatening consequences; urgent intervention, intubation, or ventilatory support indicated | Death |
| Definition: A disorder characteriz<br>with an increase in arterial levels | red by impaired gas exchange by t<br>s of carbon dioxide. | he respiratory system resulting in | hypoxemia and a decrease in oxy | genation of the tissues that may be | e associate |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight<br>gain; intervention with fluid<br>restriction and/or diuretics<br>indicated | Moderate signs or symptoms; steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; ventilatory support indicated | Death |
| Definition: A disorder characteriz retinoic acid. | zed by weight gain, dyspnea, pleur | al and pericardial effusions, leukoo | cytosis and/or renal failure original | ly described in patients treated wit | h all-trans |
| Sinus disorder | Asymptomatic mucosal crusting; blood-tinged secretions | Symptomatic stenosis or<br>edema/narrowing interfering<br>with airflow; limiting instrumental<br>ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by involvement of the paranasa | al sinuses. | • | | |
| Sleep apnea | Snoring and nocturnal sleep arousal without apneic periods | Moderate apnea and oxygen<br>desaturation; excessive daytime<br>sleepiness; medical evaluation<br>indicated; limiting instrumental<br>ADL | Oxygen desaturation;<br>associated with hypertension;<br>medical intervention indicated;<br>limiting self care ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | red by cessation of breathing for sh | nort periods during sleep. | • | ' | • |
| Sneezing | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by the involuntary expulsion of | air from the nose. | | ' | ' |
| Sore throat | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | - | - |
| Definition: A disorder characteriz | red by of marked discomfort in the | throat | • | | |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characteriz | red by a high pitched breathing sou | und due to laryngeal or upper airw | ay obstruction. | | |
| Tracheal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the trachea and another | organ or anatomic site. | | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe pain; hemorrhage or respiratory symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ted by an inflammation involving th | | | I | I_ |
| Tracheal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Stridor or respiratory distress<br>limiting self care ADL;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | red by a narrowing of the trachea. | 1 | • | • | • |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Voice alteration | Mild or intermittent change from normal voice | Moderate or persistent change<br>from normal voice; still<br>understandable | Severe voice changes including predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology | - | - |
| Definition: A disorder characteriz | ed by a change in the sound and/o | or speed of the voice. | | | |
| Wheezing | Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe respiratory symptoms<br>limiting self care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a high-pitched, whistling sou | ind during breathing. It results from | n the narrowing or obstruction of t | he respiratory airways. | |
| Respiratory, thoracic and mediastinal disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Alopecia | Hair loss of <50% of normal for | Hair loss of >=50% normal for | = | = | - |
| | that individual that is not | that individual that is readily | | | |
| | obvious from a distance but only | '' | | | |
| | on close inspection; a different | piece is necessary if the patient | | | |
| | hair style may be required to | desires to completely | | | |
| | cover the hair loss but it does | camouflage the hair loss; | | | |
| | not require a wig or hair piece to | associated with psychosocial | | | |
| | camouflage | impact | | | |
| Definition: A disorder character | ized by a decrease in density of hair | compared to normal for a given i | ndividual at a given age and body | location. | |
| Body odor | Mild odor; physician intervention | Pronounced odor; psychosocial | - | - | - |
| | not indicated; self care | impact; patient seeks medical | | | |
| | interventions | intervention | | | |
| Definition: A disorder character | ized by an abnormal body smell res | ulting from the growth of bacteria | on the body. | I | |
| Bullous dermatitis | Asymptomatic; blisters covering | Blisters covering 10 - 30% BSA; | Blisters covering >30% BSA; | Blisters covering >30% BSA; | Death |
| | <10% BSA | painful blisters; limiting | limiting self care ADL | associated with fluid or | |
| | 1.570 5571 | instrumental ADL | | electrolyte abnormalities; ICU | |
| | | illistrumental ADL | | care or burn unit indicated | |
| Definition: A diserder sharester | <br> | restorized by the presence of bull | <br> | care or barr arm maleated | 1 |
| | ized by inflammation of the skin cha | | | | |
| Dry skin | Covering <10% BSA and no | Covering 10 - 30% BSA and | Covering >30% BSA and | - | - |
| | associated erythema or pruritus | associated with erythema or | associated with pruritus; limiting | | |
| | | pruritus; limiting instrumental | self care ADL | | |
| | | ADL | | | |
| Definition: A disorder character | zed by flaky and dull skin; the pores | are generally fine, the texture is | a papery thin texture. | Ī | 1 |
| Erythema multiforme | Target lesions covering <10% | Target lesions covering 10 - | Target lesions covering >30% | Target lesions covering >30% | Death |
| | BSA and not associated with | 30% BSA and associated with | BSA and associated with oral or | BSA; associated with fluid or | |
| | skin tenderness | skin tenderness | genital erosions | electrolyte abnormalities; ICU | |
| | | | | care or burn unit indicated | |
| Definition: A disorder character | ized by target lesions (a pink-red rin | g around a pale center). | | | |
| Erythroderma | - | Erythema covering >90% BSA | Erythema covering >90% BSA | Erythema covering >90% BSA | Death |
| | | without associated symptoms; | with associated symptoms (e.g., | with associated fluid or | |
| | | | 1 | electrolyte abnormalities; ICU | |
| | | Himiting instrumental ADL | i bruntus or tenderness), ilmiund | | |
| | | limiting instrumental ADL | pruritus or tenderness); limiting self care ADL | l | |
| Definition: A disorder character | ized by generalized inflammatory er | | self care ADL | care or burn unit indicated | |
| | ized by generalized inflammatory er | ythema and exfoliation. The inflan | self care ADL nmatory process involves > 90% of | care or burn unit indicated | <br> |
| Definition: A disorder character<br>Fat atrophy | Covering <10% BSA and | ythema and exfoliation. The inflan | self care ADL nmatory process involves > 90% o Covering >30% BSA; | care or burn unit indicated | - |
| | | ythema and exfoliation. The inflan<br>Covering 10 - 30% BSA and<br>associated with erythema or | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or | care or burn unit indicated | <br> - |
| | Covering <10% BSA and | ythema and exfoliation. The inflan<br>Covering 10 - 30% BSA and<br>associated with erythema or<br>tenderness; limiting instrumental | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | <br> -<br> |
| Fat atrophy | Covering <10% BSA and asymptomatic | ythema and exfoliation. The inflan<br>Covering 10 - 30% BSA and<br>associated with erythema or | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. | ythema and exfoliation. The inflan<br>Covering 10 - 30% BSA and<br>associated with erythema or<br>tenderness; limiting instrumental<br>ADL | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, | ythema and exfoliation. The inflan<br>Covering 10 - 30% BSA and<br>associated with erythema or<br>tenderness; limiting instrumental<br>ADL | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a | ythema and exfoliation. The inflan Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient | ythema and exfoliation. The inflan Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by | ythema and exfoliation. The inflan Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or | ythema and exfoliation. The inflan Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by | ythema and exfoliation. The inflant Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or | ythema and exfoliation. The inflan Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy<br>Definition: A disorder characteri | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or | ythema and exfoliation. The inflant Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care | care or burn unit indicated | - |
| Fat atrophy Definition: A disorder characteri Hirsutism Definition: A disorder characteri | Covering <10% BSA and asymptomatic Ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | ythema and exfoliation. The inflant Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care ADL | care or burn unit indicated f the body surface area. - | and under |
| Fat atrophy Definition: A disorder characteri Hirsutism Definition: A disorder characteri | Covering <10% BSA and asymptomatic Ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | ythema and exfoliation. The inflant Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | self care ADL matory process involves > 90% of Covering > 30% BSA; associated with erythema or tenderness; limiting self-care ADL s where growth is considered to be | care or burn unit indicated f the body surface area. - | and under |
| Fat atrophy Definition: A disorder characteri Hirsutism Definition: A disorder characteri androgen control (beard, moust | Covering <10% BSA and asymptomatic Ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | ythema and exfoliation. The inflant Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | self care ADL matory process involves > 90% o Covering >30% BSA; associated with erythema or tenderness; limiting self-care ADL | care or burn unit indicated f the body surface area. - | - and under |
| Fat atrophy Definition: A disorder characteri Hirsutism Definition: A disorder characteri androgen control (beard, moust | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | ythema and exfoliation. The inflan Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact growth in women in anatomic site | self care ADL matory process involves > 90% of Covering > 30% BSA; associated with erythema or tenderness; limiting self-care ADL s where growth is considered to be | care or burn unit indicated f the body surface area. - | - and unde |
| Fat atrophy<br>Definition: A disorder characteri<br>Hirsutism | Covering <10% BSA and asymptomatic ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair ized by the presence of excess hair tache, chest, abdomen) Limited to one site (palms, | ythema and exfoliation. The infland Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact growth in women in anatomic site | self care ADL matory process involves > 90% of Covering > 30% BSA; associated with erythema or tenderness; limiting self-care ADL s where growth is considered to be Generalized involving sites | care or burn unit indicated f the body surface area. - | - and unde |
| Fat atrophy Definition: A disorder characteri Hirsutism Definition: A disorder characteri androgen control (beard, moust | Covering <10% BSA and asymptomatic Ized by shrinking of adipose tissue. In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair Ized by the presence of excess hair tache, chest, abdomen) Limited to one site (palms, soles, or axillae); self care | ythema and exfoliation. The inflant Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact growth in women in anatomic site Involving >1 site; patient seeks medical intervention; associated | self care ADL matory process involves > 90% of Covering > 30% BSA; associated with erythema or tenderness; limiting self-care ADL s where growth is considered to be Generalized involving sites other than palms, soles, or | care or burn unit indicated f the body surface area. - | - and unde |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | I | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or<br>density of hair that the patient is<br>either able to camouflage by<br>periodic shaving or removal of<br>hairs or is not concerned | Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) | - | - | - |
| | enough about the overgrowth to use any form of hair removal | plus/minus arms] that requires<br>frequent shaving or use of<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial | | | |
| Dofinition: A disorder characteri | Zod by hair dansity or langth bayon | impact | a particular body ragion for a part | icular ago or race | ļ |
| Hypohidrosis | zed by hair density or length beyon | Symptomatic; limiting instrumental ADL | Increase in body temperature; | Heat stroke | Death |
| Definition: A disorder characteri | zed by reduced sweating. | | | <b>.</b> | |
| Lipohypertrophy | Asymptomatic and covering <10% BSA | Covering 10 - 30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% BSA and<br>associated tenderness and<br>narcotics or NSAIDs indicated;<br>lipohypertrophy; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri | zed by hypertrophy of the subcutan | eous adipose tissue at the site of | multiple subcutaneous injections of | of insulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by a change in the color of the | nail plate. | T | Τ | 1 |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the<br>nail bed from the nail plate or<br>nail loss; limiting instrumental<br>ADL | - | - | - |
| Definition: A disorder characteri | zed by loss of all or a portion of the | nail. | | | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by vertical or horizontal ridges | on the nails. | ' | ' | |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensation | n in the skin. | T | Γ | 1 |
| Palmar-plantar<br>erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling, blisters, bleeding, edema, or hyperkeratosis) with pain; limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | - | - |
| | zed by redness, marked discomfort | | | reet. | Т |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by swelling due to an excessive | e accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Painless erythema and<br>erythema covering <10% BSA | Tender erythema covering 10 - 30% BSA | Erythema covering >30% BSA<br>and erythema with blistering;<br>photosensitivity; oral<br>corticosteroid therapy indicated;<br>pain control indicated (e.g.,<br>narcotics or NSAIDs) | Life-threatening consequences; urgent intervention indicated | Death |

| | Skin and subcutaneous tissue disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | T |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated;<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | - | - |
| Definition: A disorder character | ized by an intense itching sensation | | 1 | I | ' |
| Purpura | Combined area of lesions covering <10% BSA | Combined area of lesions covering 10 - 30% BSA; bleeding with trauma | Combined area of lesions covering >30% BSA; spontaneous bleeding | -<br>Dider lesions are usually a darker | -<br>purple color |
| and eventually become a browr | | | | , | |
| Rash acneiform | Papules and/or pustules<br>covering <10% BSA, which may<br>or may not be associated with<br>symptoms of pruritus or<br>tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder character | ized by an eruption of papules and p | ,<br>oustules, typically appearing in fac | ce, scalp, upper chest and back. | ' | • |
| Rash maculo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering<br>>30% BSA with or without<br>associated symptoms; limiting<br>self care ADL | - | - |
| | ized by the presence of macules (fla<br>upper trunk, spreading centripetally | | nown as morbillform rash, it is one | of the most common cutaneous a | dverse |
| Scalp pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensation | n in the skin covering the top and | the back of the head. | Γ | |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA; associated with ulceration | - | - |
| Definition: A disorder character | ized by the degeneration and thinning | ng of the epidermis and dermis. | _ | T | |
| Skin hyperpigmentation | Hyperpigmentation covering <10% BSA; no psychosocial impact | Hyperpigmentation covering >10% BSA; associated psychosocial impact | - | - | - |
| Definition: A disorder character | ized by darkening of the skin due to | excessive melanin deposition. | | | |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | - | - | - |
| Definition: A disorder character | ized by loss of skin pigment. | | | | |
| Skin induration | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| | ized by an area of hardness in the s | | T | T | |
| Skin ulceration | Combined area of ulcers <1 cm;<br>nonblanchable erythema of<br>intact skin with associated | Combined area of ulcers 1 - 2 cm; partial thickness skin loss involving skin or subcutaneous | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to or necrosis of | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or | Death |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | - | - | Skin sloughing covering <10%<br>BSA with associated signs (e.g.,<br>erythema, purpura, epidermal<br>detachment and mucous<br>membrane detachment) | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment) | Death |
| Definition: A disorder characterize mucous membranes. | ed by less than 10% total body ski | n area separation of dermis. The | syndrome is thought to be a hyper | rsensitivity complex affecting the s | kin and the |
| Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | - | - | - |
| Definition: A disorder characterize | ed by local dilatation of small vess | els resulting in red discoloration o | f the skin or mucous membranes. | 1 | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characterize mucous membranes. | ed by greater than 30% total body | skin area separation of dermis. T | he syndrome is thought to be a hy | persensitivity complex affecting th | e skin and the |
| Urticaria | Urticarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 - 30% BSA; oral intervention indicated | Urticarial lesions covering >30%<br>BSA; IV intervention indicated | - | - |
| Definition: A disorder characterize | ed by an itchy skin eruption charac | cterized by wheals with pale interio | ors and well-defined red margins. | | |
| Skin and subcutaneous tissue disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Social circumstances | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 1 2 3 4 | | | |
| Menopause | Menopause occurring at age 46 | Menopause occurring at age 40 | Menopause occurring before | - | - |
| | - 53 years of age | - 45 years of age | age 40 years of age | | |
| Definition: A disorder characteriz | ed by the permanent cessation of | menses, usually defined by 12 co | nsecutive months of amenorrhea i | n a woman over 45 years of age. | |
| Social circumstances - Other, | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | | | disabling; limiting self care ADL | | |

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| procedures - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| I | | | disabling; limiting self care ADL | | |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by leakage of intravascular flui<br>ck syndromes, low-flow states, ische | · | • | • | |
| Flushing | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Symptomatic, associated with hypotension and/or tachycardia; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by episodic reddening of the fa | ice. | i | 1 | |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a localized collection of bloo | od, usually clotted, in an organ, sp | ace, or tissue, due to a break in th | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by an uncomfortable and temp | orary sensation of intense body w | armth, flushing, sometimes accom | panied by sweating upon cooling. | |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic<br>BP 140 - 159 mm Hg or<br>diastolic BP 90 - 99 mm Hg);<br>medical intervention indicated;<br>recurrent or persistent (>=24<br>hrrs); symptomatic increase by<br>>20 mm Hg (diastolic) or to<br>>140/90 mm Hg if previously | Stage 2 hypertension (systolic<br>BP >=160 mm Hg or diastolic<br>BP >=100 mm Hg); medical<br>intervention indicated; more<br>than one drug or more intensive<br>therapy than previously used<br>indicated<br>Pediatric: Same as adult | Life-threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit, hypertensive<br>crisis); urgent intervention<br>indicated<br>Pediatric: Same as adult | Death |
| Definition: A disorder characte | rized by a pathological increase in b | WNL; monotherapy indicated<br>Pediatric: recurrent or persistent<br>(>=24 hrs) BP >ULN;<br>monotherapy indicated | | ng 140 over 90 mm Hg. | |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention or hospitalization indicated | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a blood pressure that is belo | ow the normal expected for an ind | ividual in a given environment. | | |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by the loss of lymph fluid into t | he surrounding tissue or body cav | ity. | 1 | |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery skin texture; papillary formation; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by excessive fluid collection in | tissues that causes swelling. | | | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characte | erized by a cystic lesion containing ly | mph. | 1 | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of ischemia managed non-<br>surgically and without permanent deficit | Recurring or prolonged (>=24<br>hrs) and/or invasive intervention<br>indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by impaired circulation to an ex | ktremity. | 1 | | |
| Phlebitis | - | Present | - | - | - |
| Definition: A disorder characte | rized by inflammation of the wall of a | vein. | | | |
| Superficial thrombophlebitis | - | Present | - | - | - |
| Definition: A disorder characte | erized by a blood clot and inflammation | on involving a superficial vein of th | e extremities. | | |

| | Vascular disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery) | Death |
| Definition: A disorder characteriz cough, orthopnea and headache | ed by obstruction of the blood flow | in the superior vena cava. Signs | and symptoms include swelling ar | nd cyanosis of the face, neck, and | upper arms, |
| Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | Thrombosis (e.g., uncomplicated pulmonary embolism [venous], non-embolic cardiac mural [arterial] thrombus), medical intervention indicated | Life-threatening (e.g., pulmonary embolism, cerebrovascular event, arterial insufficiency); hemodynamic or neurologic instability; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream. | <b>.</b> | |
| Vasculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the w | rall of a vessel. | • | • | |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of ischemia managed medically and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a decrease in blood supply | due to narrowing or blockage of a | visceral (mesenteric) artery. | | |
| Vascular disorders - Other, specify | 1 , 1 , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |







NIH Publication No. 09-5410 Revised June 2010 Reprinted June 2010



## APPENDIX 2. PEMPHIGUS DISEASE AREA INDEX (PDAI)

## Pemphigus Disease Area Index (PDAI)

| Skin | Activity | | Damage |
|---|---|---|---|
| Anatomical Locatio | Erosion/Blisters or new erythema | | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion |
| | absent 1-3 lesions, up to one >2 cm in any diameter, none > 6 cm 2-3 lesions, at least two > 2 cm diameter, none > 6 cm 3 lesions, none > 6 cm diameter 3 lesions, none > 6 cm diameter 3 lesions, and/or at least one >6 cm 3 lesions, and/or at least one lesion >16 cm diameter or entire area | Number<br>lesions if<br>≤ 3 | 0 absent<br>1 present |
| Ears | | | |
| Nose | | | |
| Rest of the face | | | |
| Neck | | | 00 |
| Chest | | | |
| Abdomen | | | |
| Back, buttocks | | | |
| Arms | | | 12 |
| Hands | | | 4 |
| Legs | | | |
| Feet | | | |
| Genitals | | | |
| Total skin | /120 | | /12 |
| Scalp | , | | |
| Scalp | Erosion/Blisters or new erythema | | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion<br>0 absent |
| | 0 absent 1 in one quadrant 2 two quadrants 3 three quadrants 4 affects whole skull 10 at least one lesion > 6 cm | | 1 present |
| Total Scalp (0-10) | /10 | | /1 |
| Mucous mer | nbrane | | 915 |
| Anatomical<br>Location | Erosion/Blisters | | |
| | 0 absent<br>1 1 lesion<br>2 2-3 lesions<br>5 >3 lesions or 2 lesions >2 cm<br>10 entire area | Number<br>lesions<br>if ≤ 3 | |
| Eyes | | | |
| Nose | | | |
| Buccal mucosa | | | |
| Hard palate | | | |
| Soft palate | | | |
| Upper gingiva | | | |
| Lower gingiva | | | |
| Tongue | | | |
| Floor of mouth | | | |
| Labial bucosa | | | |
| Posterior pharynx | | | |
| Anogenital | | | |
| Total Mucosa | /120 | | |

Copyright ©2007 University of Pennsylvania; All Rights Reserved.

# APPENDIX 3. AUTOIMMUNE BULLOUS DISEASE QUALITY OF LIFE (ABQOL) QUESTIONNAIRE

 Syntimmune, Inc.

## **ABQOL Questionnaire**

| Name: | Date: |
|---|---|
| DOB: Sex: M/F | Contact Number: |
| Pemphigus Subtype: Pemphigus Vulgaris | <ul> <li>Epidermolysis Bullosa Aquisita</li> </ul> |
| □ Bullous Pemphigoid | □ Linear IgA Bullous Dermatoses |
| □ Pemphigus Follaceus | □ Mucous Membrane Pemphigoid |
| □ Other | · |
| The following questions ask about the ways in quality of life. | which <i>blistering disease treatments</i> affect your |
| Please choose an option from the right hand co felt within the last week. | olumn which most closely correlates to how you |
| Please time your survey in minutes and se | conds – start time AM/PM |
| <ol> <li>In regards to your blistering disease,<br/>does your skin burn, sting or hurt in</li> </ol> | All the time Sometimes |
| any way? | Occasionally Not at all |
| 2. In regards to your blistering disease, | All the time |
| does your skin itch? | <ul><li>Sometimes</li><li>Occasionally</li></ul> |
| | Not at all |
| Have you had to change your clothing because of your blictoring | I have to be very careful with how tight my elething is and what materials they |
| clothing because of your blistering disease? | my clothing is and what materials they<br>are made of – I have had to change what<br>I wear all the time |
| | I have had to change most of the things I wear |
| | I have had to change some of the things I wear |
| | I have never had to change what I wear |
| 4. Do you notice your skin heals slowly? | I notice this all the time I notice this sometimes |
| | I notice this occasionally |
| Do you have difficulty bathing or | |
| showering because of your blistering | o Sometimes |
| disease? | Occasionally Not at all |

| In regards to your blistering disease,<br>does your mouth have erosions<br>which are painful? | <ul><li>All the time</li><li>Sometimes</li><li>Occasionally</li><li>Not at all</li></ul> |
|---|---|
| In regards to your blistering disease, do your gums bleed easily? | <ul><li> All the time</li><li> Sometimes</li><li> Occasionally</li><li> Not at all</li></ul> |
| Does your blistering disease results in you having to avoid food or drinks that you enjoy? | I can no longer eat any of the foods I used to enjoy I can eat some of the foods I enjoy I can eat most of the foods I enjoy I can eat anything I like |
| 9. As a result of your blistering disease, are you embarrassed about your appearance? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 10. Do you feel depressed or angry because of your blistering disease? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 11. Do you feel anxious or cannot relax as a result of your blistering disease? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 12. Do you worry that friends and family find your blistering skin condition tiresome? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 13. Is your blistering disease causing sexual difficulties? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 14. Does your blistering disease affect relationships with friends or loved ones? | <ul> <li>I have had to end a relationship because of my disease OR I cannot have a relationship because of my disease</li> <li>Relationships are very difficult</li> <li>Relationships are a little difficult</li> <li>This has not affected my relationships</li> </ul> |

| 15. Does your blistering disease affect your social life? | <ul> <li>I cannot go out to socialize any more</li> <li>I can only go to some social events</li> <li>I can go to most social events</li> <li>My social life is not affected</li> </ul> |
|---|---|
| 16. Does your blistering disease affect your work or study? | <ul> <li>Yes, I can no longer work or study</li> <li>Yes, I find it difficult to work or study</li> <li>Yes, it is a little harder than before to work or study</li> <li>No, I am not affected OR not applicable (N/A)</li> </ul> |
| 17. Do employers discriminate against you because of your blistering disease? | <ul> <li>I cannot find a job due to my blistering disease</li> <li>I have had to change jobs due to my blistering disease</li> <li>I still have my job but it is more difficult than before</li> <li>My employers are completely understanding OR not applicable (N/A)</li> </ul> |

Please indicate the time taken to finish the survery: minutes seconds

Thank you for taking the time to complete this questionnaire

### APPENDIX 4. SKINDEX-29

 Syntimmune, Inc.

## **DERMATOLOGY SURVEY**

This survey concerns the skin condition which has bothered you the most during the past four weeks.

These questions concern your feelings over the past 4 weeks about **the skin condition that has bothered you the most**. Check the answer that comes closest to the way you have been feeling.

| HOW OFTEN DURING THE PAST FOUR WEEKS DO THESE STATEMENTS DESCRIBE YOU? | NEVER | RARELY | SOMETIMES | OFTEN | ALL THE |
|---|---|---|---|---|---|
| 1. My skin hurts | 1 | $\square_2$ | Пз | □4 | □5 |
| 2. My skin condition affects how well I sleep | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 3. I worry that my skin condition may be serious | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 4. My skin condition makes it hard to work or do hobbies | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 5. My skin condition affects my social life | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 6. My skin condition makes me feel depressed | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 7. My skin condition burns or stings | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 8. I tend to stay at home because of my skin condition | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 9. I worry about getting scars from my skin condition | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 10. My skin itches | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 11. My skin condition affects how close I can be with those I love . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 12. I am ashamed of my skin condition | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 13. I worry that my skin condition may get worse | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 14. I tend to do things by myself because of my skin condition . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 15. I am angry about my skin condition | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 16. Water bothers my skin condition (bathing, washing hands) . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 17. My skin condition makes showing affection difficult | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 18. I worry about side-effects from skin medications / treatments . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 19. My skin is irritated | □1 | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 20. My skin condition affects my interactions with others | □1 | $\square_2$ | $\square_3$ | $\square_4$ | □5 |

Please turn to next page

These questions concern your feelings over the past 4 week about **the skin condition that has bothered you the most**. Check the answer that comes closest to the way you have been feeling.

| HOW OFTEN DURING THE PAST 4 WEEK<br>DO THESE STATEMENTS DESCRIBE YOU? | NEVER | RARELY | SOMETIMES | OFTEN | ALL THE<br>TIME |
|---|---|---|---|---|---|
| 21. I am embarrassed by my skin condition | <b>□</b> 1 | $\square_2$ | Пз | □4 | □5 |
| 22. My skin condition is a problem for the people I love | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 23. I am frustrated by my skin condition | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 24. My skin is sensitive | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 25. My skin condition affects my desire to be with people | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 26. I am humiliated by my skin condition | □1 | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 27. My skin condition bleeds | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 28. I am annoyed by my skin condition | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 29. My skin condition interferes with my sex life | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 30. My skin condition makes me tired | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |

## PROTOCOL AMENDMENT **SUMMARY OF CHANGES**

**Protocol Title:** Phase 1b/2 Multicenter, Open-Label, Safety, and Dose-Finding Study

of SYNT001 in Subjects with Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**Study Drug:** SYNT001

Syntimmune, Inc. **Sponsor:** 

116 Huntington Avenue

Suite 301

Boston, MA 02116

**Medical Monitor:** 

Wallace House

17-21 Maxwell Place Stirling, Scotland FK81JU

Mobile Phone: PPD

Office Phone: PPD

ext. PPD

**Original Protocol** 18 January 2017 1.0 21 March 2017 12 April 2017 2.0 10 October 2017 3.0 08 June 2018 4.0

#### CONFIDENTIALITY STATEMENT

This document is the property of Syntimmune, Inc. This document contains confidential information, which should not be copied, referred to, released, or published without written approval from Syntimmune. Investigators are cautioned that the information given in this brochure might be subject to change and revision. Any conclusion regarding efficacy and safety must be considered provisional.

Version 4.0

#### BACKGROUND

Protocol amendment Version 4.0 of the SYNT001-103 protocol was issued on 07 June 2018.

Since the design of the original protocol, the Sponsor has completed longer SYNT001 nonclinical toxicology studies (14-weeks vs 5-weeks). Additionally, the Sponsor has gained experience with conducting the trial and has learned about logistical issues affecting the successful execution of the protocol to obtain preliminary safety and effectiveness data.

For a number of reasons, including inclusion and exclusion criteria, prohibited and permitted medications, and logistical burden of study conduct (eg, number and complexity of study visits), enrollment into study SYNT001-103 has been far slower than anticipated. Further, as currently designed, the study will provide only limited information on dose selection to support further clinical development (eg, duration of dosing and potential role of a loading dose approach cannot be assessed). Preliminary safety results support good safety and tolerability of SYNT001 at 10 mg/kg for 5 weekly doses. Regarding efficacy, data thus far support proof-of-concept for SYNT001 in pemphigus; however, it appears that longer dosing will be needed to maintain response and higher doses may lead to a higher response rate and robustness of response.

Syntimmune therefore is amending the SYNT001-103 protocol to address the above issues. The Study Assessments have been extensively modified to decrease the complexity of the study and make the execution of the study more acceptable to potential subjects and more feasible for study sites; changes include the removal of 7 study visits and organization of study visits into major and minor visits with more consistent assessments. It is anticipated that these changes should facilitate study enrollment, especially when combined with additional adjustments to the inclusion and exclusion criteria and prohibited medications, including removal of the upper limit on body mass index (previously was 39.9 kg/m<sup>2</sup>) and allowance for steroid tapering prior to screening. To better inform dose selection and pivotal trial design, dosing in Cohort 3 has been extended from 5 weekly doses to 14, and an optional Cohort 4 has been added to allow exploration of an alternate dose level (maximum of 45 mg/kg) and dosing duration (up to 14 weekly doses) to be determined following data review by the Dose Escalation Committee (DEC). This option could include a loading dose followed by lower weekly doses. To gain more information on dose selection, endpoints regarding extent of lowering of total IgG levels and change in the Pemphigus Disease Area Index (PDAI) total activity score from baseline have been added as a primary objective in addition to safety.

Administrative changes in the amendment include changes in the medical monitor and Sponsor contact information. General grammatical, typographical, and formatting updates have been made throughout the document to provide consistency and clarity, reduce redundancy, and improve readability.

### **SUMMARY OF CHANGES**

With this update, the following changes since Version 3.0 have been made:

 Table 1.
 Summary of Changes: Protocol Version 4.0

| Section<br>Number and<br>Title | Description of Change |
|---|---|
| Cover Page | Protocol Title |
| | • Revised to indicate updated Phase 1b/2 status and dose finding intent to commence under Cohorts 2, 3, and optional Cohort 4. |
| | • Removed tolerability as a quantifiable measurement as the focus of the trial will be safety. |
| | <ul> <li>Medical term for primary indication revised from chronic pemphigus to<br/>pemphigus to more closely reflect eligibility criteria and terminology<br/>commonly used by treating physicians.</li> </ul> |
| | Other |
| | • The Medical Monitor's title and Syntimmune Inc. address have been updated for accuracy. |
| Section 1,<br>Protocol<br>Synopsis | The protocol synopsis has been modified to more closely align with industry standards and the National Institute of Health (NIH)/Food and Drug Administration (FDA) protocol template. Below is a summary of changes; refer to the changes described for the individual protocol sections for more detail: |
| | Added the sponsor, Syntimmune Inc. |
| | • Indicated the company's intentions to open study sites outside the United States of America to support subject enrollment. |
| | • The study rationale is now an overview of protocol Section 2, Background and Rationale. |
| | • Study objectives have been grouped with study endpoints; study objectives now only appear once in the protocol synopsis. |
| | <ul> <li>The study design not only describes changes to cohorts but now<br/>includes the role of the Dose Escalation Committee (DEC) and<br/>stopping and dose escalation rules.</li> </ul> |
| | • Study methodology has been separated from study design and is now in a stand-alone section. |
| | • The inclusion and exclusion criteria have been modified as described in Section 6 Study Population. |
| | <ul> <li>Additional detail has been added to Duration of subject participation<br/>and Study drug, dosage, and administration.</li> </ul> |
| | • Prohibited Concomitant treatments has now been changed to Permitted and Prohibited Concomitant Treatments. |

| | • The following sections have been removed from the synopsis, but content remains in the protocol text to reduce redundancy: |
|---|---|
| | <ul> <li>Safety assessments</li> </ul> |
| | o Pharmacokinetics |
| | o Pharmacodynamics/Activity |
| | o Immunogenicity |
| | <ul> <li>Skin biopsy</li> </ul> |
| | o Photography |
| | • In the statistical consideration section, the intent to treat (ITT) study population has been changed to Safety population. Analyses have been updated to reflect additional detail included in the study endpoints. |
| | <ul> <li>Subheadings have been added to clearly delineated content.</li> </ul> |
| Study Diagram | Study Diagram has been added changing the dose, number of doses and timing of DEC reviews for Cohorts 2 and 3 and adding optional Cohort 4 to reflect changes to study design. |
| | • Cohort 1 number of subjects has been modified from 8 to up to 8. |
| | • Cohort 2 dose has been modified to ≤30 mg/kg and the number of subjects reduced from 8 to 4. |
| | • Cohort 3 has been added with ≤ 30 mg/kg and number of doses extended to 14 in 4 subjects. |
| | • The optional cohort has shifted from Cohort 3 to 4 with a maximum dose of 45 mg/kg and maximum number of doses out to 14. |
| | • Timing of DEC data reviews for Cohorts 2 and 3 is after 50% of subjects reach Day 42. |
| | • The DEC may now lower the dose within a cohort and add up to 4 additional patients to Cohorts 2, 3, and optional Cohort 4. |
| Schedule of | Table 3 (Cohort 2) |
| Events | • Efforts were made to simplify the study of events to reduce subject and site burden and increase flexibility with visit scheduling, as described below: |
| | <ul> <li>A total of 7 visits have been removed (Days 1, 2, 5, 12, 19, 29, and 20).</li> </ul> |
| | <ul> <li>Day 33 has been changed to Day 35 to shift to a weekly visit<br/>schedule out to 1 month after the final dose.</li> </ul> |
| | <ul> <li>Visit windows have been increased as outlined below:</li> </ul> |
| | <ul><li>Weekly visits: ± 1 day</li></ul> |
| | ■ Every other week visit: ± 3 days |
| | ■ Monthly visits: ± 5 days |
| | • Specific changes to the Schedule of Events as compared to Cohort 1 (Table 2) are described below. Many of the changes support |

categorization of Treatment and Follow-up visits into major and minor visits. All minor visits have the same schedule of testing. Tests conducted at major visits are now more consistent.

- Pemphigus Disease Area Index (PDAI), physical examination, and anti-desmoglein (1 and 3) antibody titers are being done at every visit.
- Tetanus and Varicella Zoster testing will now be done at set timepoints (Baseline, Day 56, and Day 112).
- Pharmacokinetic (PK) sampling will only be done at Baseline and the day of the final SYNT001 final dose.
- o Immunogenicity is no longer done at Day 84.
- Testing of biomarkers has been reduced [complement component 3 (C3), anti-epithelial cell antibody (AECA), RNAseq, urine immunoglobulin G (IgG), and immunophenotyping]. These biomarkers are now only done at Baseline, Day 35, and Day 56.
- o Photography is no longer done at Day 14 and Day 84.
- o Added Health-related Quality of Life (HR-QoL) questionnaires to Baseline, Day 35, Day 56, and Day 112.

#### Table 4 (Cohort 3)

- Assessments done at Screening, Baseline and Follow-up visits align with Cohort 2 (Table 3).
- Treatment will extend from 5 to 14 doses and subjects will receive weekly IV infusions during this time.
  - Assessments at the mid-point of dosing and the final dose (major visits) align with Cohort 2 (Table 3).
  - Assessments at all other treatment visits (minor visits) also align with Cohort 2 (Table 3).

## Table of Contents

The overall structure of the document has been modified slightly to improve readability and usability:

- Study Objectives and Endpoints have been logically grouped together under Section 3.0.
- Study Drug section has been moved up in the protocol due to its importance and now falls directly after Study Objectives and Endpoints. The content has not fundamentally changed but has been organized into recognizable sections for easy reference.
- The order of Study Procedures in Section 7 now more closely reflects the Schedule of Events.
- A section has been added for HR-QoL questonnaires to mirror the updated Schedule of Events.
- Study Assessments section now details Cohort 2 Schedule of Events and the extended dosing out to 14 doses for Cohort 3.

| | Section 9 title has been changed from Removing Subjects from Study to Study Rules. Lost to Follow-up was added as a sub-section. |
|---|---|
| | • The Safety section has been reorganized for improved readability and now includes the Procedures in Case of Emergency that was previously at the start of the document. |
| | • Vaccinations, Management of Allergic or Infusion Reactions, and Potential Immune Effects are grouped under Warnings and Precautions (Section 10.3). |
| | • Overdose has been added to Other Safety Considerations (Section 10.5). |
| | • Multiple sections were collapsed into 1 comprehensive section titled Study Management (Section 12). |
| | Tables have been added to reflect the new study design and assessments by cohort. |
| | • Appendices have been added for the new HR-QoL questionnaires, the Autoimmune Bullous Disease Quality of Life (ABQoL) and Skindex-29. |
| | Figure 1 was added to illustrate the study design. |
| List of<br>Abbreviations | The table was updated to include all abbreviations throughout the synopsis and protocol text. Each abbreviation was defined the first time used in both the synopsis and protocol text. |
| Section 2, | Background and Rationale |
| Background and Rationale | • Text has been added to describe SYNT001's predicted mechanism of action. |
| | Additional indications identified as IgG-mediated autoimmune disorders have been added. |
| | Study Rationale |
| | The study rationale has been updated to include dose activity criteria and remove tolerability criteria. |
| | Selection of Doses in this Study |
| | Non-human primate (NHP) data is now described before the healthy volunteer study (Phase 1a) to follow the chronology of when the studies completed. Information about the completed 14-week toxicology study has been added. |
| Section 3, Study | Study objectives and endpoints have not fundamentally changed but |
| Objectives and | have been rewritten to more closely align with industry standards. |
| Endpoints | An objective and endpoint have been added for dose selection to define pritorio to select a dose for future eliminal testing. |
| | <ul> <li>criteria to select a dose for future clinical testing.</li> <li>Edits have been made to ensure each objective has a corresponding</li> </ul> |
| | endpoint and vice versa. |

| | A 11 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
|---|---|
| | An objective and endpoint have been added for the HR-QoL guestiannaires; the HR QoL will be used to better understand the |
| | questionnaires; the HR-QoL will be used to better understand the subject experience when being dosed with SYNT001. |
| Section 4, Study | Description of SYNT001 |
| Drug | <ul> <li>Windows for the SYNT001 infusion duration (±15 minutes) have been</li> </ul> |
| Drug | added to account for procedural and patient differences. |
| | Dose Requirements |
| | It has been clarified that subject doses will be limited to 5000 mg. A |
| | subject with a body weight that extrapolates to a dose > 5000 mg, will |
| | only receive 5000 mg. |
| Section 5, Study | The study design has been updated to reflect changes in dose, number of |
| Design | doses and timing of DEC reviews for Cohorts 2 and 3 and adding optional |
| | Cohort 4. |
| | • Cohort 1 number of subjects modified from 8 to <u>up to</u> 8. |
| | • Cohort 2 dose modified to $\leq$ 30 mg/kg and reduced the number of |
| | subjects from 8 to 4. |
| | • Cohort 3 has been added with $\leq$ 30 mg/kg and number of doses to 14 in |
| | 4 subjects. |
| | • The optional cohort has shifted from Cohort 3 to 4 with a maximum |
| | dose of 45 mg/kg and maximum doses out to 14. |
| | • Timing of DEC Data Reviews for Cohorts 2 and 3 is after 50% of |
| | subjects reach Day 42. |
| | • The DEC may now lower the dose within a cohort and add up to 4 |
| | additional patients in to Cohorts 2, 3, and optional Cohort 4. |
| | Study Rules were not included, as done in the corresponding synopsis |
| | section; instead Section 9 (Study Rules) is referenced. |
| Section 6, Study | Target Population |
| Population | Based on the new study design, the total number of subjects has been |
| | updated to 20 with a possible additional 12 subjects pending DEC |
| | evaluation. |
| | o Enrollment into Cohort 2 onwards revised from 8 to 4 subjects |
| | with an additional optional 4 subjects per cohort pending DEC |
| | evaluation. Inclusion Criteria |
| | <ul> <li>#4b. Expanded list of concomitant immunosuppressants to include</li> </ul> |
| | methotrexate, dapsone, cyclosporine, tacrolimus, sirolimus, |
| | cyclophosphamide. Parameter of stable dose raised from <10% to |
| | <25% change in dose and window narrowed from 6 weeks to 4 weeks |
| | prior to screening. |
| | • #4c. Change in dose of concomitant corticosteroids considered |
| | acceptable during the 2 weeks prior to screening changed from a 10% |
| | change in dose to an increase in dose by 50%. |

- #4d. Expanded list of allowable topical therapies for pemphigus lesions to include low-strength hydrocortisone (≤ 1%), tacrolimus, sirolimus, pimecrolimus, and dexamethasone elixir solution.
- #4e. If not on regular corticosteroids, no pulse corticosteroids are allowed in the 2 weeks prior to screening.
- #5. Eliminated upper body mass index (BMI) limit of 39.9 kg/m<sup>2</sup>.
- #10. Added a PDAI total severity score of >4 at screening.

#### **Exclusion Criteria**

- #6. Reduced intravenous immunoglobulin (IVIG) treatment window prior to screening from 60 days to 30 days.
- #9. Reduced plasmapheresis or immunoadsorption treatment window prior to screening from 60 to 30 days.
- #11. Clarified that systemic or topical immunosuppressive drugs are excluded unless specified in the inclusion criteria.

#### Section 7, Study Procedures

- Pulse oximetry has been included under vital sign measurements.
- Table 6 with timing windows for PK/pharmacodynamic (PD) Sampling, electrocardiogram (ECG), and Vital Sign Measure has been moved to the Study Procedures Section.
  - The timing windows for Cohorts 2, 3, and optional Cohort 4 were added.
  - Windows were separated from the pharmacokinetic sampling windows.
- RR Interval as a required part of the ECG assessments has been added back into the protocol.
- Blood volumes for clinical laboratory measurements have been recalculated to align with changes to the Schedule of Events.
- Serum tetanus antibody and varicella-zoster virus antibody testing has been simplified and will be done at set timepoints.
- For Cohorts 2, 3, and optional Cohort 4, PK parameters studied will be maximum plasma concentration determined directly from the concentration-time profile (C<sub>max</sub>) and observed time to reach peak plasma concentration (T<sub>max</sub>).
- Pharmacodynamic Assessment (Table 8) has been updated to include timing of testing for Cohorts 2 and 3.
- Clarified that immunogenicity testing will also include determination of anti-drug antibody (ADA) titer.
- Section for HR-QoL questionnaires has been added to mirror the updated Schedule of Events.
- Optional skin biopsies will not be collected after Cohort 1.

### **Prior and Concomitant Medications**

 Reordered and relocated language under newly created subsection headers, Permitted Medications and Prohibited Medications. Key changes include:

Permitted Medications

• #5. Use of medication to treat infusion reactions.

| Section 9, Study<br>Rules | <ul> <li>#6. Low-strength corticosteroids applied to a single lesion.</li> <li>#7. Topical tacrolimus, sirolimus or pimecrolimus applied to a single lesion.</li> <li>#8. Dexamethasone elixir solution for oral lesions.</li> <li>#9. Stable use of immunosuppressants: tacrolimus, sirolimus, pimecrolimus, methotrexate, cyclophosphamide, and dapsone.</li> <li>#10. One month after the final dose of SYNT001, corticosteroids may be tapered at the Investigator's discretion.</li> <li>Prohibited Medications</li> <li>#4. IV corticosteroids prior to infusion (except in subjects who received corticosteroids for treatment of a prior infusion reaction to SYNT001).</li> <li>#7. Vaccinations post treatment window reduced from 56 days to 28 days.</li> <li>Deleted corticosteroid taper instructions.</li> <li>Subject Withdrawal</li> <li>Subjects that require a significant increase in dose(s) of anti-pemphigus medications(s) for the management of their pemphigus will be encouraged to return for follow-up visits to capture safety data.</li> <li>Dose Escalation Stopping Rule</li> <li>The description of dose escalation stopping rules now reflects the new</li> </ul> |
|---|---|
| | <ul><li>study design.</li><li>The DEC now has the ability to reduce the dose within a cohort and</li></ul> |
| | potentially add study subjects to a given cohort. |
| Section 10,<br>Evaluation of<br>Safety | The content of this section has not changed substantially, but text has been reorganized to improve flow and ability to locate critical information in the case of a safety event. |
| Section 11,<br>Statistical<br>Considerations | <ul> <li>General design has been updated to mirror the protocol title.</li> <li>Dose selection data will be evaluated based on IgG response and PDAI score reduction.</li> <li>Study drug serum concentrations will be calculated by C<sub>max</sub> and T<sub>max</sub> for Cohorts 2, 3 and optional Cohort 4.</li> </ul> |
| Section 12,<br>Study<br>Management | <ul> <li>Study Administrative Structure table has been updated with Medical Director and a new Sponsor Contact information.</li> <li>Informed Consent procedures have been edited to add International Council on Harmonisation Good Clinical Practice (ICH GCP) compliance language.</li> <li>Subject confidentiality and privacy language have been added to clarify Health Insurance Portability and Accountability Act (HIPPA) confidentiality guarantees and data protection.</li> <li>Audits and inspections may be performed by the sponsor to ensure validity of study data.</li> </ul> |
| Global Changes | Edits and formatting changes have been made throughout to improve clarity and readability. |
- Typographical and formatting corrections as well as corrections for consistency have been made.
- Renamed sections and subsections to reflect content and protocol naming conventions. Reordered language under modified or newly created subsection headers.
- Consolidated language if repeated in more than one section of protocol.
- Naming convention for sponsor changed from Syntimmune to Sponsor.
- Chronic pemphigus revised to pemphigus to indicate accepted medical terminology.
- Nomenclature for investigational product revised to study drug for consistency.
- Medical Monitoring and Sponsor contact information updated.

# SYNTIMMUNE, INC. CLINICAL STUDY PROTOCOL

A Phase 1b/2, Multicenter, Open-Label, Safety, and Dose-Finding Study of SYNT001 in Subjects with Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

IND Number: 132727 Study Drug: SYNT001

**Sponsor:** Syntimmune, Inc.

116 Huntington Avenue

Suite 301

Boston, MA 02116

**Medical Monitor:** PF

Wallace House

17-21 Maxwell Place Stirling, Scotland FK81JU

Mobile Phone: PPD Office Phone: PPD

ext. PPD

 Original Protocol:
 18 January 2017

 Amendment 1.1:
 21 March 2017

 Amendment 2.0
 12 April 2017

 Amendment 3.0
 10 October 2017

 Amendment 4.0
 08 June 2018

 Amendment 5.0
 18 September 2018

#### CONFIDENTIALITY STATEMENT

The information contained herein is confidential and the proprietary property of Syntimmune, Inc. Any unauthorized use or disclosure of such information without the prior written authorization of Syntimmune is expressly prohibited.

## SPONSOR SIGNATURE

I have read and approve this protocol. My signature, in conjunction with the signature of the Investigator, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Guideline for Good Clinical Practice (GCP), the United States Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| PPD | |
|----------------|-------------------|
| | 19 SEPT 2018 |
| | Date of Signature |
| Syntimmune Inc | |

#### **INVESTIGATOR SIGNATURE**

I have read and approve this protocol. My signature, in conjunction with the signature of the Sponsor, confirms the agreement of both parties that the clinical study will be conducted in accordance with the protocol and all applicable laws and regulations including, but not limited to, the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Guideline for Good Clinical Practice (GCP), the United States Code of Federal Regulations (CFR), and the ethical principles that have their origins in the Declaration of Helsinki.

| Nothing in this document is intended to lim | it the authority of a physicia | n to provide emergency |
|---|---|---|
| medical care under applicable regulations. | | |

| Investigator Signature | Date of Signature |
|-------------------------------------|-------------------|
| Name of Investigator (please print) | <del></del> |

# 1. SYNOPSIS

| Study title | A Phase 1b/2, Multicenter, Open-Label, Safety, and Dose-Finding Study of |
|---|---|
| | SYNT001 in Subjects with Pemphigus (Vulgaris or Foliaceus) |
| Sponsor | Syntimmune, Inc. |
| Protocol number | SYNT001-103 |
| Clinical phase | Phase 1b/2 |
| Number of study centers | Approximately 20 global study sites |
| Study rationale | Pemphigus is a potentially life-threatening group of rare blistering autoimmune diseases that affect the skin and mucous membranes. The exact cause is unknown, though autoantibodies are thought to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. The prognosis of pemphigus has markedly improved over the last decades with steroid therapy. Nevertheless, mortality remains an issue (1.6% to 12% of cases) (Hsu et al., 2016; Kasperkiewicz et al., 2017; Langan et al., 2008). In these cases, death typically occurs as a consequence of treatment-related systemic infections and in a smaller proportion, as a consequence of superinfected lesions. While steroids have greatly improved patient outcomes, they are associated with serious and long-lasting side effects; therefore, their use should be limited as much as possible. Although other currently available treatments for certain autoimmune disorders, including immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 monoclonal antibodies (mAbs), such as rituximab, can be effective, they can be associated with significant adverse effects and delayed or non-durable responses. SYNT001 targets key mechanisms contributing to pathology in a variety of immunoglobulin G (IgG)-mediated autoimmune disorders. When administered to healthy subjects, SYNT001 has been shown to significantly decrease total IgG, as well as immune complexes with which IgG is associated. Based on these results, it is predicted that SYNT001 will also reduce the levels of pathogenic autoantibodies. This could lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce circulating immune complexes (CICs) and the associated innate and adaptive immune responses may allow for sustained disease modification. Thus, this study is being conducted to evaluate the safety and |
| | modification. Thus, this study is being conducted to evaluate the safety and immunogenicity and determine a minimally effective dose (MED) of intravenous (IV) SYNT001 in pemphigus patients. |

| Study objectives and endpoints | The study objectives and their corresponding endpoints (primary, secondary, and exploratory) are detailed below. | |
|---|---|---|
| | <b>Primary Objectives</b> | Primary Endpoints |
| | Safety: To evaluate the safety of IV infusions of SYNT001 at different dose levels and dosing regimens in subjects with pemphigus (vulgaris or foliaceus) | Safety: The evaluation of SYNT001 safety based on vital signs, physical examinations, electrocardiograms (ECGs), clinical safety laboratory tests, the incidence of adverse events (AEs), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) summarized by dose and dosing regimen, severity, and relationship to study drug |
| | Dose Selection: To determine a MED of SYNT001 as assessed by (i) total IgG level nadir and (ii) the proportion of subjects that meet the criteria for response by Pemphigus Disease Area Index total activity score (PDAI) | Dose Selection: The determination of dose and dosing regimen of SYNT001 that achieves (i) total IgG level nadir decrease by ≥60% and ≤90% from baseline and (ii) a PDAI total activity score of ≥50% reduction from baseline to allow further clinical development in subjects with pemphigus (vulgaris or foliaceus) |
| | Secondary Objectives | Secondary Endpoints |
| | To evaluate the efficacy of doses of SYNT001 at different dose levels and dosing regimens on pharmacodynamics (PD) biomarkers | The evaluation of PD biomarkers based on absolute serum levels and percent change from baseline of total IgG, IgG subtypes (IgG1-4), immunoglobulin A (IgA), immunoglobulin M (IgM), albumin, and CIC summarized by dose, dosing regimen and visit |

| To determine the pharmacokinetics (PK) of SYNT001 following IV infusions at different dose levels and dosing regimens | The determination of PK parameters including half-life (t <sub>1/2</sub> ), maximum serum concentration determined directly from the concentration-time profile (C <sub>max</sub> ), observed time of peak serum concentration (T <sub>max</sub> ), area under the serum concentration-time curve from pre-dose (time <sub>0</sub> ) to 24 hours post-dose (AUC <sub>0-24</sub> ), and area under the serum concentration-time curve from pre-dose (time <sub>0</sub> ) to infinity (AUC <sub>0-∞</sub> ), (Cohort 1); maximum serum concentration determined directly from the maximum serum concentration and corresponding T <sub>max</sub> (Cohort 2) summarized by dose, dosing regimen, visit and time point |
|---|---|
| To assess the efficacy of doses of SYNT001 at different dose levels and dosing regimens on disease markers | <ul> <li>The assessment of pemphigus disease activity by responses on the PDAI based on absolute and percent change from baseline, summarized by dose, dosing regimen and visit</li> <li>The assessment of pemphigus disease activity by pathogenic antibody levels based on absolute and percent change from baseline of serum antidesmoglein 1 and 3 antibody (anti-Dsg 1 and anti-Dsg 3) levels summarized by dose, dosing regimen and visit</li> </ul> |
| To measure the immunogenicity of SYNT001 administered at different dose levels and dosing regimens | The immunogenicity of SYNT001 as determined by presence of anti-SYNT001 binding antibodies and neutralizing antibodies summarized by dose, dosing regimen, visit and time point |
| <b>Exploratory Objectives</b> | <b>Exploratory Endpoints</b> |
| To explore the effect of SYNT001 at different dose levels and dosing regimens on biomarkers to understand the pathophysiology of the disease and the SYNT001 mechanisms of action | The exploration of SYNT001 mechanisms of action and effects of SYNT001 on pathophysiology summarized by dose, dosing regimen and visit as determined by: |

| To determine the impact of different SYNT001 dose levels and dosing regimens on the subject's use of corticosteroids to treat their | <ul> <li>Complement component 3 levels by nephelometry</li> <li>Anti-epithelial cell antibody (AECA) titers by indirect immunofluorescence</li> <li>Fc gamma R2A receptor (FCGR2A) single nucleotide polymorphisms (SNP) by genotyping</li> <li>Presence of disease and inflammatory markers by total RNA sequencing</li> <li>Immunophenotyping including measurements of T cells, monocytes, natural killer (NK) cells and B cells by flow cytometry</li> <li>Urine IgG levels to explore SYNT001 distribution and elimination (Cohort 1 only)</li> <li>Exploratory biomarkers to investigate immune response associated with pemphigus</li> <li>The evaluation of corticosteroid use during the study will be summarized by dose, dosing regimen and visit</li> </ul> |
|---|---|
| pemphigus (vulgaris or foliaceus) To assess the impact of SYNT001 on the subject's health-related quality of life (HR-QoL) at different dose levels and dosing regimens | The assessment of SYNT001 impact on subject's health-related quality of life (HR-QoL) by responses to the Autoimmune Bullous Diseases Quality of Life (ABQoL) questionnaire and Skindex-29 scores summarized by dose, dosing regimen and visit |
| To assess the effect of SYNT001 on<br>the appearance of skin and mucosal<br>lesions at different dose levels and<br>dosing regimens | The qualitative assessment of changes in appearance of skin and mucosal lesions as determined by photography presented by dose, dosing regimen and visit |
| To quantify the amount of SYNT001 in skin (skin biopsies optional) | The determination of SYNT001 levels in skin biopsies across timepoints (skin biopsies optional) (Cohort 1 only) |

#### Study design

This is a multicenter, open-label safety study to determine the dose regimen of SYNT001 administered IV in subjects with pemphigus (vulgaris or foliaceus).

Up to 8 subjects with a diagnosis of pemphigus (vulgaris or foliaceus) will receive SYNT001 10 mg/kg weekly x 5 doses (Cohort 1).

Up to 12 subjects with a diagnosis of pemphigus (vulgaris or foliaceus) will receive SYNT001 30 mg/kg weekly x 3 doses (Loading), followed by SYNT001 10 mg/kg every other week x 5 doses (Maintenance) (Cohort 2).

Subjects in both cohorts will complete the following periods of assessment: Screening, Treatment, and Follow-Up. For Cohort 1 details of the dosing schedule and assessments, see Table 2. For Cohort 2 details, see Table 3.

The Dose Escalation Committee (DEC) will consist of the Medical Monitor, an Independent Clinical Expert and the Sponsor Medical Lead. The DEC may request that Investigators, other experts, or members within their organization participate in the review. Additional information on the DEC's responsibilities is provided in Section 9.5 and the DEC Charter.

An overview of the study cohorts is provided in Table 1 and Figure 1 shows a schematic of the study design.

| 7D 11 4 | <b>~</b> 1 | · |
|----------|------------|----------|
| Table 1. | Cohort ( | Overview |

| Cohort<br>No. | No. of<br>Subjects | SYNT001<br>Dose | No. of<br>Doses | Frequency of Doses |
|---|---|---|---|---|
| 1ª | Up to 8 | 10 mg/kg | 5 | Weekly |
| 2 <sup>b</sup> | Up to 12 | Loading:<br>30 mg/kg <sup>c</sup> | 3° | Weekly <sup>c</sup> |
| | | Maintenance:<br>10 mg/kg <sup>c</sup> | 5° | Every other week <sup>c, d</sup> |

- a. No more than 3 subjects with pemphigus foliaceus may be enrolled
- b. Two or fewer subjects with pemphigus foliaceus may be enrolled
- c. The dose, number of doses, and frequency of doses in Cohort 2 will be confirmed based on review of safety and PD evaluations, including but not limited to, dose-limiting toxicities, AEs, TEAEs, SAEs, and total IgG levels. Following Sponsor review of emerging safety, PD and efficacy data, the Loading dose may be reduced to 20 or 10 mg/kg weekly and/or the Maintenance dose may be increased to 20 or 30 mg/kg every other week and/or dose frequency may be increased to weekly.
- d. Ongoing safety and PD evaluations may result in modification of the dose and dosing regimen in Cohort 2. See APPENDIX 5 for the corresponding visit schedule.

Subjects will be enrolled at staggered intervals to facilitate adequate safety evaluation before dosing of subsequent subjects .

At 24-hour and 7-day intervals described below, all available safety data (including but not limited to dose limiting toxicities [DLTs], AEs, TEAEs, SAEs and PD (including but not limited to total IgG levels), will be reviewed.

#### Safety Review of 24-hour Data for Cohorts 1 and 2, Subject 1

• The first 2 subjects in each cohort will be dosed at least 24 hours apart. A DEC review of the 24-hour safety data for the first subject in Cohort 1 will be performed to ensure that there are no overt safety concerns

| | before dosing the second subject. The Sponsor Medical Lead and Medical Monitor will conduct the 24-hour safety data review for the first subject in Cohort 2. |
|---|---|
| | Safety Review of 7-day Data for Cohorts 1 and 2, Subjects 1 and 2 |
| | • The 7-day safety data for the first 2 subjects in Cohort 1 will be reviewed by the DEC prior to dosing the remaining subjects in the cohort. The Sponsor Medical Lead and Medical Monitor will conduct the 7-day safety data review in Cohort 2. |
| | The 24-hour and 7-day reviews will consider seriousness and severity of AEs/TEAEs/SAEs and relatedness to study drug, vital sign assessments, physical examinations, and clinical laboratory testing. |
| | Safety data (including but not limited to DLTs, AEs, TEAEs, SAEs), and PD data (including but not limited to IgG levels) will be reviewed on an ongoing basis by the Medical Monitor and the Sponsor Medical Lead. In addition, at any point the DEC may initiate a review of all cumulative data if requested by a DEC member. |
| | <ul> <li>If a DLT occurs, dosing will be halted within that cohort and dose-escalation will not occur. NOTE: DLTs will be defined generally as severe (Grade 3) AEs occurring in ≥2 subjects that are determined to be clinically significant and considered related to study drug.</li> <li>If any subject at any time during the study experiences a life-threatening AE (Grade 4) that is considered related to study drug, further dosing in all enrolled subjects will be suspended.</li> <li>At any time during the study, the study or any ongoing study cohort may be discontinued if the Sponsor Medical Lead determines that further drug exposure would pose an undue risk to subjects.</li> </ul> |
| | Dosing for any individual subject will be discontinued (ie, no further administration of SYNT001) if the subject experiences any study drug-related SAE or any study drug-related non-serious AE that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired), or in the judgement of the Sponsor Medical Lead, suggests that it could be unsafe to administer further study drug to that subject. |
| Number of subjects | Up to 20 subjects are planned; up to 8 subjects in Cohort 1 and up to 12 subjects in Cohort 2. Subjects who withdraw for any reason other than an AE may be replaced. |
| Study population | Male or female subjects 18 years of age and older with a confirmed diagnosis of pemphigus (vulgaris or foliaceus) |
| Diagnosis and main | Inclusion criteria: |
| entry criteria | Subjects must meet the following criteria to be eligible for the study: |
| | <ol> <li>Willing and able to read, understand, and sign an informed consent form.</li> <li>Male or female ≥18 years of age at the time of screening.</li> <li>Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:</li> </ol> |

- a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/or skin lesions).
- b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal (ULN).
- c. History of at least one positive tissue-based test (eg, biopsy, direct immunofluorescence [DIF]).
- 4. Active disease defined as lesions lasting >2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion >1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 mAb, last dose >9 months prior to screening.
  - b. If being treated with other immunosuppressants (ie, azathioprine, mycophenolate mofetil, methotrexate, dapsone, cyclosporine, tacrolimus, sirolimus, or low-dose cyclophosphamide [≤100 mg/day]), dose must be stable, defined as <25% change in dose, for 4 weeks prior to screening.</li>
  - c. On stable dose of corticosteroids, defined as ≤1 mg/kg of prednisone or equivalent and may not be increased by more than 50% in the 2 weeks prior to screening.
  - d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth.
  - e. Stable use of topical low strength hydrocortisone (≤1%), tacrolimus, sirolimus, or pimecrolimus for lesions contributing <10% of the PDAI total activity score for the 4 weeks prior to screening is allowed. Stable use of dexamethasone elixir solution (swish and spit only) for oral lesions for the 4 weeks prior to screening is allowed.
  - f. If not on regular corticosteroids, no pulse corticosteroids are allowed in the 2 weeks prior to screening.
- 5. Body mass index (BMI)  $> 18.5 \text{ kg/m}^2$ .
- 6. Has a negative pregnancy test documented prior to the first dose of study drug (for women of childbearing potential).
- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the screening period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through the final study visit.
- 10. A PDAI total activity score of >4 at screening.

#### **Exclusion criteria:**

Subjects meeting any of the following criteria are ineligible for the study:

- 1. Subject unable or unwilling to comply with the protocol.
- 2. Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ).
- 3. Positive for human immunodeficiency virus (HIV) or hepatitis C antibody.
- 4. Positive for hepatitis B surface antigen.
- 5. Active infection or history of recurrent infections.
- 6. IVIG treatment within 30 days of screening.
- 7. Received any cytotoxic (other than azathioprine) or any non-anti-CD20 mAb therapy in the 3 months prior to screening.
- 8. Any exposure to an investigational drug or device within the 30 days prior to screening.
- 9. Plasmapheresis or immunoadsorption within 30 days of screening.
- 10. Cellular therapy, including chimeric antigen receptor and T-cell (CAR-T), at any time prior to screening.
- 11. Use of any systemic or topical immunosuppressive drugs within 3 months of screening not including those allowed by the inclusion criteria.
- 12. Serum total IgG <600 mg/dL at screening.
- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (eg, a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results).
- 14. Any vaccination within 2 weeks of screening.

# Study drug, dosage, and administration

#### **Study drug:** SYNT001

#### **Dosages:**

Cohort 1: 10 mg/kg x 5 weekly doses

Cohort 2: 30 mg/kg x 3 weekly doses (Loading) followed by 10 mg/kg every other week x 5 doses (Maintenance).

The dose, number of doses, and frequency of doses in Cohort 2 will be confirmed based on ongoing review of safety and PD evaluations, including but not limited to, DLTs, AEs, TEAEs, SAEs, and total IgG levels. Following Sponsor review of emerging safety, tolerability, PD and efficacy data, the Loading dose may be reduced to 20 or 10 mg/kg weekly and/or the Maintenance dose may be increased to 20 or 30 mg/kg every other week and/or dose frequency may be increased to weekly.

#### **Product presentation and preparation:**

SYNT001 provided as a liquid at a nominal concentration of 50 mg/mL. SYNT001 is diluted in dextrose 5% in water (D5W) to prepare the solution for infusion.

**Route of administration:** IV in 250 mL over 1 hour  $\pm$  15 minutes Investigators may adjust the duration of the infusion if needed to improve tolerability.

| Control doss and | Not applicable | | | | | |
|---|---|---|---|---|---|---|
| Control, dose, and route of | Not applicab | ole . | | | | |
| administration | | | | | | |
| Duration of subject | The duration | of subject pa | rticipation for | r each cohort | is as follows | s: |
| participation | Cohort Screening Treatment Follow-up Maximum Total | | | | | |
| | | | | | Days | Weeks |
| | 1 | ≤14 days | 28 days | 84 days | 126 days | 18 weeks |
| | 2 | ≤14 days | 84 days | 56 days | 154 days | 22 weeks |
| | | 1 | I . | | II. | |
| Permitted and prohibited concomitant treatments | All pemphigus treatments a subject receives within at least 3 months prior to enrollment and all other treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented. Permitted Medications | | | | | |
| | Concomitant | medication a | and treatment | for co-existing | ng conditions | s, including |
| | | | permitted if no | | | |
| | <ol> <li>Topical</li> <li>Topical</li> <li>Concome experien</li> <li>Medication acetamir (eg, rani)</li> <li>Low-stressingle le</li> <li>Topical contribut</li> <li>Dexame throughout</li> <li>Stable reazathiop cyclospocyclopho</li> </ol> | or systemic tradidocaine for the didocaine for the didocaine for the didocaine for the didocaine for potent headache: the didocaine, famotic ength topical discontributed acrolimus, since the sone elixing the sone elixing trial partice of the gimen of the rine, mycophorine, tacrolimus psphamide (\lequip exphamide) | e study. ial infusion-re ial infusion-re ial infusion-re ial infusion-re ial infusion-re ial infusion, diphe<br>dine). corticosteroid ing <10% of rolimus or pir the PDAI tota solution for c ipation (swish following systemolate mofet ius, sirolimus 100 mg/day). | oral candidia<br>relief as nee<br>cally indicate<br>elated reaction<br>may recommenhydramine<br>s (eg, hydrocothe PDAI tothe<br>mecrolimus and activity seconal lesions it<br>in and spit only<br>temic immunial, low-dose in conticostero | sis. ded. ed for any AF ens (IRRs), in nend prophyl , histamine <sub>2</sub> ( cortisone ≤1% al activity sc pplied to a si ore. To dose remain ly). nosuppressan methotrexate ids, or low defined. | Es the subject cluding post-actic use of (H <sub>2</sub> ) blockers 6) applied to a ore. ngle lesion as stable ats: , dapsone, ose oral |
| | at the Investi | Fourteen days after the final dose of SYNT001, corticosteroids may be tapered at the Investigator's discretion. | | | | |
| | Prohibited I | | | | | |
| | | ollowing medi<br>ove as permitt | | ot be permit | ted during the | e study unless |
| | <ul><li>2. Monocle</li><li>3. Any topi</li><li>are listee</li><li>4. IV cortice</li><li>corticost</li></ul> | onal antibodie<br>cal or system<br>l as permitted<br>costeroids pric | or to infusion atment of a pr | tudy drug<br>opressive dru<br>(except in su | bjects who re | eceived |

6. Vaccinations within 2 weeks of screening through 28 days following final dose of study drug

#### **Corticosteroids**

#### Before enrollment

The dose of corticosteroids taken for pemphigus or any other condition prior to screening must be at a dose  $\leq 1$  mg/kg and the dose level must have not increased in dose level by more than 50% in the 2 weeks prior to screening. No pulse dosing of steroids is permitted in the 2 weeks prior to screening.

#### From screening until 2 weeks after the last dose of SYNT001

The dose of corticosteroids taken for pemphigus or any other condition should remain stable (<10% change in dose level) from screening until 2 weeks after the last dose of SYNT001. Corticosteroids should neither be started nor discontinued during this period with the exception of subjects who experience an IRR that requires corticosteroids as part of the management of the IRR. Such subjects may receive corticosteroids prophylactically prior to subsequent SYNT001 infusions at the discretion of the Investigator.

# From 2 weeks after the last dose of SYNT001 until end of study participation

At the discretion of the Investigator, but only after at least 2 weeks beyond the last dose of SYNT001, a slow corticosteroid taper may be started as per the following suggested schedule:

• If on >30 mg of prednisone per day, decrease by no more than 10 mg every two weeks until a final dose.

If per the Investigator's judgement, the subject would benefit from a change to the pemphigus treatment beyond the allowed steroid taper, this will be considered on a case-by-case basis in consultation with the Sponsor.

# Statistical considerations

Three populations will be employed in the analysis of study data:

- The Safety population will consist of all subjects who have received at least one dose of study drug.
- The PD population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.
- The PK population will consist of all subjects who receive at least one dose of study drug and have post-dose PK data available.

Primary safety analyses will be performed on the safety population. Demographics, subject disposition, screening, and baseline characteristics will be summarized for the Safety, PD and PK populations, where appropriate.

#### Sample size

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

#### Criteria for evaluation

Baseline analysis

Baseline characteristics to include medical history, physical examination, vital signs, and ECG will be summarized using descriptive statistics by dose, dose regimen, and visit.

#### Safety analysis

The evaluation of SYNT001 based on vital signs, physical examination, ECGs, clinical safety laboratory tests, the incidence of AEs, TEAEs, and SAEs summarized by dose and dose regimen, severity, and relationship to study drug.

#### Dose-finding analysis

The evaluation of SYNT001 based on total IgG levels and responses on the PDAI total activity score from baseline will be summarized using descriptive statistics by dose and dose regimen, visit and time point, as applicable.

#### Statistical methodology

Treatment-emergent AEs (TEAEs) will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least one occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study drug [related/not related]) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject and dose using SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by time point, dose, and dose regimen. The incidence of laboratory abnormalities will be summarized. The worst onstudy grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, or above the normal limits of the central laboratory. Vital sign measurements and change from baseline will be summarized at each scheduled time point using descriptive statistics. PD/PK results will be summarized by dose and dosing regimen. Descriptive statistics of PD/PK parameters for SYNT001 will include mean, standard deviation (SD), coefficient of variation (CV), median, minimum, and maximum.

Immunogenicity results will be summarized by cohort, visit and time point. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

Disease activity marker results will be summarized by dose, dose regimen, and visit. Descriptive statistics will include mean, SD, median, minimum, and maximum.

PDAI results will be summarized by score (total activity score, total damage score), cohort, and visit. Descriptive statistics will include absolute change from baseline and percent change from baseline.

Additional statistical analyses may be performed.

Figure 1. Cohort Enrollment



**Table 2.** Study Assessments for Cohort 1

| | Screening | | | | | | | Tre | atment | Period | | | | | | | Follo | w-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 |
| Time point (study day) | -14 to -1 | 0 | 1 | 2 | 5 <sup>p</sup> | 7 | 12 <sup>p</sup> | 14 | 19 <sup>p</sup> | 21 | 28 | 29 | 30 | 33 | 42 | 56 | 84 | 112 or |
| | | | (±1 h) | (±2 h) | (±4 h) | (±6 h) | (±6 h) | (±6 h) | (±6 h) | (±6 h) | (±6 h) | (±1 h) | (±2 h) | (±4 h) | (±3 d) | (±5 d) | (±5 d) | ET (±5 d) |
| Informed consent | X | | | | | | | | | | | | | | | | | |
| Demographics/medical history | X | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | | | | | | | | |
| Physical examination <sup>a</sup> | X | X | | | | X | | X | | X | X | | | | X | X | X | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>c</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Clinical safety labs <sup>d</sup> | X | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | | | | | | | | | | | | X | | X |
| Hepatitis and HIV screen | X | | | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>f</sup> | X | X | | | | | X | | | | X | | | | | X | | |
| Tetanus and VZV antibodies <sup>g</sup> | | X | | | | | | | | | | | | | | X | X | X |
| PDAI | | X | | | | X | | X | | X | X | | | X | X | X | X | X |
| PK sampling <sup>h</sup> | | X | X | X | X | | | | | | X | X | X | X | | | | |
| Immunogenicity <sup>i</sup> | | X | | | | | | X | | | X | | | | | X | X | X |
| Study drug administration <sup>j</sup> | | X | | | | X | | X | | X | X | | | | | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4) <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Xq |
| CIC | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Anti-Dsg (1 and 3) antibody titers | X | X | | | | X | | X | | | | | | X | | X | X | X |
| C3 and AECA <sup>1</sup> | | X | | | | | | X | | | | | | X | | X | X | X |
| FCGR2A by buccal swab <sup>m</sup> | | X | | | | | | | | | | | | | | | | |
| RNAseq | | X | | | | | | X | | | | | | X | | X | X | X |
| Urine IgG | | X | | | | | | X | | | | | | X | | X | X | X |
| Immunophenotyping <sup>n</sup> | | X | | | | | | | | | X | | | | | X | | |
| Exploratory pemphigus immune response biomarkers | | X | | | X | X | X | X | X | X | X | | | X | X | X | X | X |
| Optional skin biopsy | | X | X | X | | | | X | | | | | | X | | X | X | |
| Photography <sup>o</sup> | | X | | | | | | | | | | | | X | | X | X | X |
| Adverse events | | | | | To be co | ollected | from the | e date th | at the IC | CF is sig | ned thro | ugh the | last stud | ly visit | | | | |
| Concomitant medications | | | | | | | | ithin 14 | | | | | | | | | | |

Abbreviations: CIC = circulating immune complexes; d = days; ECG = electrocardiogram; ET = early termination; h = hour(s); HIV = human immunodeficiency virus; ICF = informed consent form; PDAI = Pemphigus Disease Area Index; PK = pharmacokinetic; VZV = varicella zoster virus.

- a. Complete physical examination, including weight, to be performed. Height and BMI will be additional assessments conducted at screening.
- b. **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. On Days 0, 7, 14, 21, and 28, vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour, and 2 hours following completion of the infusion.
- c. **Pulse oximetry:** On Days 0, 7, 14, 21, and 28, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- d. Clinical safety labs: hematology, clinical chemistry, and urinalysis (see Section 7.5 for a complete list). Full clinical safety laboratory draws will be collected at screening and on Days 0, 7, 14, 21, 28, 33, 42, 56, 84, and 112.
- e. **Pregnancy test (women of childbearing potential only):** To be performed at time of screening, prior to first dose of SYNT001 on Day 0, and on Days 56 and 112. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.
- f. Digital 12-lead ECG to be obtained in triplicate at least 1 to 2 minutes apart and after 5 minutes of rest in a supine position. See Section 7.6 for additional information. On Days 0 and 28 to be obtained 5 minutes after the completion of infusion. Day 12 ECG will be collected only if the visit is conducted at the study site.
- g. **Serology**: Testing at Day 56 will not be done for any subject whose baseline titer is below the level of detection. If the Day 56 results are greater than 30% below the baseline value, or if the subject falls below the level of detection, the subject will be re-tested at Day 84; if still below the baseline value (or level of detection), the subject will be re-tested at Day 112. Any subject whose baseline value for tetanus or VZV was above the detectable level at baseline, and is not within 30% of the baseline value or is below the detectable level by Day 112, will be referred to their primary care physician for further management. See Section 7.5.3 for additional information.
- h. **PK**: Starting on Days 0 and 28, serum samples will be collected just prior to the start of study drug infusion (pre-dose), and at 5 minutes and 2, 4, 6, 24, and 48 hours after the end-of-study drug infusion. Additional samples will be collected on Days 5 and 33. See Section 7.5.4 for additional information.
- Immunogenicity: Samples will be collected pre-dose when collected on dosing days. Samples will be collected on Days 0, 14, 28, 56, 84 and 112. See Section 7.5.6 for additional information.
- j. Prior to **study drug infusion**, SYNT001 drug product is to be diluted in dextrose 5% in water (D5W) to a total volume of 250 mL and administered intravenously over 1 hour using a 0.2-micron inline filter. See Section 4 and Section 7.8 for additional information.
- k. Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, IgM at every visit. On Days 0, 7, 14, 21, and 28, samples are collected prior to infusion of study drug. See Section 7.5.5 for additional information.
- 1. **Exploratory pharmacodynamic samples (C3 and AECA):** Collected pre-dose when collected on dosing days. See Section 7.5.5 for complete information.
- m. Buccal samples to be collected and stored; pending review of clinical and pharmacodynamics assessments.
- n. Immunophenotyping by flow cytometry for measurement of CD3+CD4+ T, CD3+CD8+ T, monocytes, NK cells and B cells.
- o. Photographs of active lesions taken prior to first dose on Day 0. Follow-up photographs will be taken at Days 33, 56, 84 and 112. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- p. Visit Days 5, 12, and 19 may be conducted via at-home nurse in lieu of a subject visit to the study site.
- q. Subjects will return to the clinic on Days 84 and 112 for follow-up visits. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 112 visit will be referred for further management.

Table 3. Study Assessment for Cohort 2

| | Screening | | Loadin | g | | | Maintenand | e | | ] | Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
| Time Point<br>(Study Day) | -14 to -1 | 0<br>Baseline | 7<br>(±1 d) | 14<br>(±1 d) | 28<br>(±3 d) | 42<br>(±3 d) | 56<br>(±3 d) | 70<br>(±3 d) | 84<br>(±3 d) | 91<br>(±5 d) or<br>ET visit | 112<br>(±5 d) | 140<br>(±5 d)<br>EOS |
| Informed consent | X | | | | | | | | | | | |
| Demographics/medical history | X | | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | | |
| Physical examination <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>c</sup> | | X | X | X | X | X | X | X | X | | | |
| Clinical safety labs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | X | | | | | X | | X |
| Hepatitis and HIV screen | X | | | | | | | | | | | |
| 12-lead ECG <sup>f</sup> | X | X | | X | X | | | | | X | | X |
| Tetanus and VZV antibodies <sup>g</sup> | | X | | | X | | | | | X | | X |
| PDAI <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| PK sampling <sup>i</sup> | | X | X | X | X | | | | X | | | |
| Immunogenicity <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Study drug administration <sup>k</sup> | | X | X | X | X | X | X | X | X | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4) <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X | $X^q$ |
| CIC | | X | X | X | X | X | X | X | X | X | X | X |
| Anti-Dsg (1 and 3) antibody titers | X | X | X | X | X | X | X | X | X | X | X | X |
| C3 and AECA <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| FCGR2A by buccal swab <sup>n</sup> | | X | | | | | | | | | | |
| RNA sequencing | | X | | | X | | | | | X | | |
| Immunophenotyping <sup>o</sup> | | X | | | X | | | | | X | | |
| Exploratory pemphigus immune response biomarkers | | X | X | X | X | X | X | X | X | X | X | X |
| Photography <sup>p</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| HR-QoL assessments | | X | | | X | | | | | X | | X |

| Adverse events | To be collected from the date that the ICF is signed through the last study visit |
|---|---|
| Concomitant medications | To be collected from within 14 days prior to Day 0 through the last study visit |

Abbreviations: CIC = circulating immune complexes; d = day(s); ECG = electrocardiogram; EOS = end of study; ET= early termination; FcGR2a= Fc gamma R2a receptor; HIV = human immunodeficiency virus; HR-QoL = health-related quality of life; ICF = informed consent form; Ig = immunoglobulin; PDAI = Pemphigus Disease Area Index; PK = pharmacokinetic; VZV = varicella-zoster virus

- a. Complete physical examination, including weight, to be performed. Height and body mass index will be additional assessments conducted at screening only.
- b. **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. Vital sign measurements will be taken on all study visits. On dosing days, vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- c. **Pulse oximetry**: On dosing days, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour, and 2 hours following completion of the infusion.
- d. Clinical safety labs: hematology, clinical chemistry, and urinalysis. See Section 7.5 for a complete list. Full clinical safety lab draws will be collected at screening and at all study visits prior to infusion if applicable.
- e. **Pregnancy test (women of childbearing potential only):** To be performed at time of screening and prior to dose on dosing days if applicable. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.
- f. Digital 12-lead ECG to be obtained after 5 minutes of rest in the supine position and in triplicate approximately 1 minute apart. See Section 7.6 for additional information. On days of treatment, to be obtained approximately 5 minutes after the completion of infusion.
- g. **Serology:** Any subject whose baseline value for tetanus or VZV was above the protective level at baseline and is not within 30% of the baseline value or is below the protective level by End of Follow-up, will be referred to their primary care physician for further management. See Section 7.5.3 for additional information.
- h. PDAI will be administered at screening. Subject eligibility requires a PDAI total activity score >4. Thereafter, assuming eligibility, the PDAI will be administered during Treatment Period and Follow-up Period. See Section 7.7 for additional information.
- i. **PK:** Starting on dosing days, serum samples will be collected just prior to the start of study drug infusion (pre-dose) and at 5 minutes, 1 and 2 hours after the end of study drug infusion. See Section 7.5.4 for additional information.
- j. Immunogenicity: Samples will be collected pre-dose when collected on dosing days. See Section 7.5.6 for additional information
- k. Prior to **study drug infusion**, SYNT001 drug product is to be diluted in dextrose 5% in water to a total volume of 250 mL and administered intravenously over 1 hour ±15 minutes using a 0.2-micron, inline filter. See Section 4 for additional information.
- 1. Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, and IgM at every visit. On dosing days, samples are collected prior to infusion of study drug. See Section 7.5.5 for additional information.
- m. Exploratory pharmacodynamic samples (C3 and AECA): Collected pre-dose when collected on dosing days. See Section 7.5.5 for complete information.
- n. Buccal samples to be collected pre-dose.
- o. **Immunophenotyping** by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, natural killer (NK) cells, and B cells. Collect samples pre-dose on dosing days.
- p. Photographs of all active lesions taken pre-dose on dosing days. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- q. Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at the Day 140 visit will be referred for further management.

# **TABLE OF CONTENTS**

| 1. | SYN | NOPSIS | 4 |
|---|---|---|---|
| LIS | ST OF | F TABLES | 24 |
| LIS | ST OF | F FIGURES | 24 |
| LIS | ST OF | F APPENDICES | 24 |
| LIS | ST OF | F ABBREVIATIONS | 25 |
| 2. | BAG | CKGROUND AND RATIONALE | 28 |
| | 2.1 | Study Rationale | 28 |
| | 2.2 | Selection of Doses in this Study | 29 |
| | 2.3 | Compliance Statement | 31 |
| 3. | STU | UDY OBJECTIVES AND ENDPOINTS | 32 |
| 4. | STU | UDY DRUG | 34 |
| | 4.1 | Description of SYNT001 | 34 |
| | 4.2 | Dose Requirements | 34 |
| | 4.3 | Handling and Storage of SYNT001 | 34 |
| | 4.4 | Study Drug Accountability | 34 |
| 5. | STU | UDY DESIGN | 35 |
| | 5.1 | Study Sites | 35 |
| | 5.2 | Overview of Study Design | 35 |
| | 5.3 | Randomization and Blinding | 36 |
| | 5.4 | Duration of Subject Participation. | 36 |
| 6. | STU | UDY POPULATION | 37 |
| | 6.1 | Target Population | 37 |
| | 6.2 | Inclusion Criteria | 37 |
| | 6.3 | Exclusion Criteria | 38 |
| 7. | STU | UDY PROCEDURES | 39 |
| | 7.1 | Informed Consent | 39 |
| | 7.2 | Demographics and Medical History | 39 |
| | 7.3 | Physical Examination. | 39 |
| | 7.4 | Vital Sign Measurements | 39 |
| | 7.5 | Clinical Laboratory Measurements | 41 |
| | 7. | 7.5.1 Pregnancy Testing | 41 |
| | 7. | 7.5.2 Virology | 42 |
| | 7. | 7.5.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody | Testing42 |
| | 7. | 7.5.4 Pharmacokinetics (PK) Sampling | 42 |
| | 7. | 7.5.5 Pharmacodynamic Sampling | 42 |
| | 7. | 7.5.6 Immunogenicity Testing | 43 |
| | 7.6 | 12-Lead Electrocardiogram (ECG) | 44 |

| | 7.7 | Pemp | phigus Disease Area Index (PDAI) | 44 |
|---|---|---|---|---|
| | 7.8 | Stud | y Drug Administration | 44 |
| | 7.9 | Photo | ographs | 44 |
| | 7.10 | Heal | th-Related Quality of Life Assessments | 44 |
| | 7.11 | Adve | erse Event Assessments | 45 |
| | 7.12 | Prior | and Concomitant Medications | 45 |
| | 7.13 | Skin | Biopsy | 47 |
| 8. | STU | DY AS | SSESSMENTS | 48 |
| | 8.1 | All C | Cohorts: Screening Period and First Treatment (Day 0) | 48 |
| | 8.1 | 1.1 | All Cohorts: Screening Period (Day -14 to Day -1) | 48 |
| | 8.1 | 1.2 | All Cohorts: Enrollment and First Treatment (Day 0) | 49 |
| | 8.2 | Coho | ort 1: Day 1 to 84 | 50 |
| | 8.2 | 2.1 | Cohort 1: Follow-up Day 1 | 50 |
| | 8.2 | 2.2 | Cohort 1: Follow-up Day 2 | 50 |
| | 8.2 | 2.3 | Cohort 1: Follow-up Day 5 | 50 |
| | 8.2 | 2.4 | Cohort 1: Treatment Day 7 (Dose 2) | 51 |
| | 8.2 | 2.5 | Cohort 1: Follow-up Day 12 | 52 |
| | 8.2 | 2.6 | Cohort 1: Treatment Day 14 (Dose 3) | 52 |
| | 8.2 | 2.7 | Cohort 1: Follow-up Day 19 | 53 |
| | 8.2 | 2.8 | Cohort 1: Treatment Day 21 (Dose 4) | 53 |
| | 8.2 | 2.9 | Cohort 1: Treatment Day 28 (Dose 5) | 54 |
| | 8.2 | 2.10 | Cohort 1: Follow-up Day 29 | 55 |
| | 8.2 | 2.11 | Cohort 1: Follow-up Day 30 | 55 |
| | 8.2 | 2.12 | Cohort 1: Follow-up Day 33 | 56 |
| | 8.2 | 2.13 | Cohort 1: Follow-up Day 42 | 56 |
| | 8.2 | 2.14 | Cohort 1: Follow-up Day 56 | 57 |
| | 8.2 | 2.15 | Cohort 1: Follow-up Day 84 | 57 |
| | 8.3 | Coho | ort 2: Subsequent Treatments to Follow-up | 58 |
| | 8.3 | 3.1 | Cohort 2: Treatment Days 7, 14, 42, 56, 70, and 84 | 58 |
| | 8.3 | 3.2 | Cohort 2: Treatment Day 28 | 59 |
| | 8.3 | 3.3 | Cohort 2: Follow-up Day 112 | 60 |
| | 8.4 | | Cohorts: End of Study or Early Termination Visit; Cohort 1, Day 11 ays 91 and 140 | |
| 9. | STU | 1 | ULES | |
| | 9.1 | | ect Withdrawal | |
| | 9.2 | • | ect Replacement | |
| | 9.3 | | y Discontinuation | |
| | 9.4 | | to Follow-up | |

| 9.5 | Stopp | ing Rules | 63 |
|---|---|---|---|
| 9. | 5.1 | Dose-Escalation Stopping Rule (Cohort 1) | 63 |
| 9. | 5.2 | Study Stopping Rule | |
| 9. | 5.3 | Individual Stopping Rule | 63 |
| 10. EVA | LUAT | ION OF SAFETY | 65 |
| 10.1 | Safety | y Parameters | 65 |
| 10.2 | Adve | rse Events | 65 |
| 10 | ).2.1 | Recording an Adverse Event | 66 |
| 10 | ).2.2 | Assessment of Causality | 66 |
| 10 | ).2.3 | Serious Adverse Events | 66 |
| | 10.2.3 | 3.1 Recording a Serious Adverse Event | 67 |
| | 10.2.3 | Reporting a Serious Adverse Event | 68 |
| 10 | ).2.4 | Follow-Up of Adverse Events and Serious Adverse Events | 69 |
| 10.3 | Warn | ings and Precautions | 69 |
| 10 | ).3.1 | Vaccinations | 69 |
| 10 | ).3.2 | Management of Allergic or Infusion-Related Reactions | 69 |
| 10 | ).3.3 | Potential Immune Effects | 73 |
| 10.4 | Event | s of Special Interest | 74 |
| 10.5 | Other | Safety Considerations | 74 |
| 10 | ).5.1 | Laboratory Data | 74 |
| 10 | ).5.2 | Medication Errors | 75 |
| 10 | ).5.3 | Overdose | 75 |
| 10 | ).5.4 | Pregnancy. | 75 |
| 11. STA | TISTIC | CAL CONSIDERATIONS | 76 |
| 11.1 | Gener | ral Design | 76 |
| 11.2 | Study | Populations | 76 |
| 11.3 | Samp | le Size Justification | 76 |
| 11.4 | Statis | tical Analysis | |
| 11 | 1.4.1 | Statistical Analysis Plan. | 76 |
| 11 | 1.4.2 | Statistical Methodology | 77 |
| 11 | 1.4.3 | Analysis of Primary Endpoints | 77 |
| | 11.4.3 | 3.1 Safety Analysis | 77 |
| | 11.4.3 | 3.2 Dose Selection Data | 78 |
| 11 | 1.4.4 | Analysis of Secondary Endpoints | 78 |
| | 11.4.4 | 4.1 Pharmacokinetic Analysis | 78 |
| | 11.4.4 | 4.2 Pharmacodynamic Analysis | 78 |
| | 11.4.4 | 1.3 Immunogenicity Analysis | 78 |
| | 11 4 4 | 1.4 PDAI Data | 78 |

| | 11 | .4.5 | Analysis of Exploratory Endpoints | 79 |
|---|---|---|---|---|
| | | 11.4. | 5.1 Corticosteroid Use | 79 |
| | | 11.4. | 5.2 Health-Related Quality of Life Data | 79 |
| | | 11.4. | 5.3 Photography | 79 |
| | 11.5 | Interi | im Analysis | 79 |
| 12. | STU | DY M | ANAGEMENT | 80 |
| | 12.1 | Regu | llatory and Ethical Considerations | 80 |
| | 12 | .1.1 | Ethical Conduct. | 80 |
| | 12 | .1.2 | Informed Consent | 80 |
| | 12 | .1.3 | Subject Confidentiality and Privacy | 80 |
| | 12 | .1.4 | Future Use of Stored Specimens | 81 |
| | 12.2 | Study | y Administration | 81 |
| | 12 | .2.1 | Institutional Review Board Approval | 82 |
| | 12 | .2.2 | Data Handling and Record Keeping | 82 |
| | 12 | .2.3 | Data Protection | 82 |
| | 12 | .2.4 | Study Site Regulatory Documentation | 82 |
| | 12 | .2.5 | Subject Clinical Source Documents and Background Data | 83 |
| | 12 | .2.6 | Electronic Case Report Forms | 84 |
| | 12.3 | Clinic | cal Monitoring, Audits, and Inspections | 84 |
| | 12 | .3.1 | Clinical Monitoring. | 84 |
| | 12 | .3.2 | Audits and Inspections | 85 |
| | 12.4 | Chan | nges to the Protocol | 85 |
| | 12.5 | Study | y Discontinuation and Closure | 85 |
| 13. | PUB | LICAT | ΓΙΟΝ AND DATA SHARING POLICY | 86 |
| 14. | REFI | EREN | CES | 87 |

# **LIST OF TABLES**

| Table 1.Cohort Overview | 8 |
|---|---|
| Table 2.Study Assessments for Cohort 1 | 16 |
| Table 3.Study Assessment for Cohort 2 | 18 |
| Table 4.Cohort Overview | 35 |
| Table 5.Timing window allowances for PK/PD sampling, ECG, and vital sign measurer at dosing visits | |
| Table 6.Clinical Safety Laboratory Panels | |
| Table 7.Pharmacodynamic Assessments | |
| Table 8.Grading and Management of Allergic or Infusion-Related Reactions | |
| Table 9.Study Administrative Structure | 82 |
| Table 10. Study Assessments for Cohort 2 (Alternate Weekly Dosing Option) | 94 |
| LIST OF FIGURES Figure 1.Cohort Enrollment | 15 |
| Figure 2.Management of Moderate (Grade 2) Infusion Reactions | |
| Figure 3.Management of Severe (Grade 3 or Higher) Infusion Reactions | |
| LIST OF APPENDICES | |
| APPENDIX 1.NCI CTCAE, Version 4.03 | 89 |
| APPENDIX 2.Pemphigus Disease Area Index (PDAI) | |
| APPENDIX 3. Autoimmune Bullous Disease Quality of Life (ABQoL) Questionnaire | 91 |
| APPENDIX 4.Skindex-29 | 92 |
| APPENDIX 5 Cohort 2 alternate schedule of events table | 93 |

#### LIST OF ABBREVIATIONS

ABQoL Autoimmune Bullous Disease Quality of Life

ADA anti-drug antibodies

AE adverse event

AECA Anti-epithelial cell antibody ALT alanine aminotransferase AST aspartate aminotransferase

AUC<sub>0-24</sub> area under the serum concentration-time curve from pre-dose (time<sub>0</sub>) to 24 hours post-

dose

AUC<sub>0-∞</sub> area under the serum concentration-time curve from pre-dose (time<sub>0</sub>) to infinity

BLQ below the limit of quantification

BMI body mass index BUN blood urea nitrogen

C1q complement component 1q C3 complement component 3

CAR-T chimeric antigen receptor and T-cell

CFR Code of Federal Regulations
CIC circulating immune complexes

C<sub>max</sub> maximum serum concentration determined directly from the concentration-time

profile

CRO contract research organization

CV coefficient of variation
D5W dextrose 5% in water
DEC Dose Escalation Committee
DIF direct immunofluorescence
DLT dose-limiting toxicity
DNA deoxyribonucleic acid

dsDNA double-stranded deoxyribonucleic acid

Dsg desmoglein

ECG electrocardiogram

eCRF electronic case report form EDC electronic data capture

eGFR estimated glomerular filtration rate

ET early termination

FCGR2A Fc gamma R2a receptor FcRn neonatal Fc receptor

FDA Food and Drug Administration

GCP Good Clinical Practice
GLP Good Laboratory Practice

H<sub>2</sub> histamine<sub>2</sub>

HBV hepatitis B virus HCV hepatitis C virus

HIPAA Health Insurance Portability and Accountability Act

HIV human immunodeficiency virus
HR-QoL health-related quality of life
IB Investigator's Brochure
IC immune complex

ICF Informed Consent Form

ICH International Council for Harmonisation of Technical Requirements for

Pharmaceuticals for Human Use

**IgA** immunoglobulin A IgG immunoglobulin G IgG1-4 immunoglobulin G1-G4 IgM immunoglobulin M **IND** investigational new drug IRB institutional review board **IRR** infusion-related reaction **IUD** Intrauterine device

IV intravenous

IVIG intravenous immunoglobulin

LDH lactate dehydrogenase
LLN lower limit of normal
mAb monoclonal antibody
MED minimum effective dose

MedDRA Medical Dictionary for Regulatory Activities

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NHP nonhuman primate NK natural killer

NOAEL no observed adverse effect level

PD pharmacodynamics

PDAI Pemphigus Disease Area Index

PK pharmacokinetic

QTcF corrected QT interval using Fridericia's formula

RNA ribonucleic acid
RNAseq RNA sequencing
SAE serious adverse event
SAP statistical analysis plan
SAS Statistical Analysis System

SD standard deviation

SNP single nucleotide polymorphism

SOC system organ class

SYNT001 a humanized, affinity matured IgG4-kappa monoclonal antibody

 $t_{1/2}$  Half-life

TEAE treatment-emergent adverse event

 $T_{max}$  observed time to reach peak plasma concentration

ULN upper limit of normal
US United States of America
VZV varicella zoster virus

WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

#### 2. BACKGROUND AND RATIONALE

SYNT001, a humanized, affinity-matured IgG4-kappa monoclonal antibody (mAb), blocks immunoglobulin G (IgG) and IgG immune complex (IC) interactions with the neonatal crystallizable fragment receptor (FcRn), and inhibits the varied roles of FcRn in the immune response.

Through specific and high affinity blockade of FcRn, SYNT001 has been shown to increase the catabolism of IgG and IgG IC in healthy volunteers and is predicted to block the ability of IgG IC to activate intracellular signaling events associated with binding to FcRn. This predicts that SYNT001 will also accelerate degradation of endogenous circulating IgG autoantibodies and IgG-IC specifically involved in the pathogenesis of autoimmunity. Blocking FcRn interactions with IgG ICs further predicts that SYNT001 will have consequences for innate and adaptive cellular immunity. In the first instance, blocking multimeric IgG IC interactions with FcRn within antigen-presenting cells should result in inhibition of IC-mediated inflammatory cytokine production and release by these cells. In addition, as FcRn determines the intracellular itinerary of IgG ICs within and among compartments important in cellular immunity, it is further anticipated that SYNT001 will block antigen processing and presentation of antigens contained within ICs that would otherwise lead to CD8<sup>+</sup> and CD4<sup>+</sup> T cell activation. Thus, SYNT001 is expected to specifically target immune functions associated with IgG and IC that are involved in certain IgG-mediated autoimmune conditions.

SYNT001 targets key mechanisms contributing to pathology in a variety of IgG-mediated autoimmune disorders.

While current treatments for certain autoimmune disorders, including chronic steroids, immunosuppressants, intravenous immunoglobulin (IVIG), plasmapheresis, and anti-CD20 mAbs, such as rituximab, can be effective, they are associated with significant adverse effects, and delayed or non-durable responses.

Pemphigus is a rare group of blistering autoimmune diseases that affect the skin and mucous membranes. Autoantibodies are thought to play an important pathogenic role in the mucosal and cutaneous manifestations in patients with pemphigus. Administration of SYNT001 significantly decreases total IgG levels, including a corresponding decrease in the levels of the pathogenic autoantibodies. This may lead to a decrease in the mucosal and cutaneous manifestations in patients with pemphigus. Moreover, the ability of SYNT001 to reduce IgG ICs and the associated innate and adaptive immune responses may allow for further sustained disease modification.

#### 2.1 Study Rationale

This study is being conducted to evaluate the safety, dose, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of intravenous (IV) SYNT001 as well as its effects on pemphigus disease activity markers.

#### 2.2 Selection of Doses in this Study

The initial SYNT001 dose levels for study SYNT001-103 were selected following careful review of the safety, tolerability, and PD effect on total IgG levels studied in non-human primates (NHP) and healthy male subjects.

Four repeat-dose toxicology studies in cynomolgus monkeys examined 2 to 14 repeat weekly IV doses 5 to 100 mg/kg SYNT001 with up to a 4-week follow-up. There was one death in the 14-week study attributed to an immune-evoked infusion reaction, which correlated with the development of anti-drug antibodies (ADAs), circulating immune complexes, circulating complement depletion, and deposition of immune complexes containing SYTN001 and complement in tissues. Across studies, clinical signs were limited to reports of transient emesis/vomitus following dosing and facial flushing and periocular swelling observed in the 5-week study after the third dose coincident with the first appearance of ADAs. With the exception of emesis/vomitus, these clinical signs were effectively controlled with diphenhydramine pretreatment in the 5-week study and the subsequent 14-week study. There were no adverse SYNT001-related changes in weight gain, clinical chemistry, gross or histo-pathology. The No Observed Adverse Effect Level (NOAEL) was the highest dose tested in all 4 studies and the overall NOAEL following repeat weekly exposure to STYNT001 of up to 14 doses in cynomolgus monkeys was 100 mg/kg.

The safety, tolerability, and PD effect on total IgG levels in study SYNT-101—a Phase 1a study that assessed single ascending doses of SYNT001 in healthy male subjects—were also reviewed. In study SYNT-101, the doses of SYNT001 up to and including 30 mg/kg were well tolerated. There were no dose-limiting toxicities, serious adverse events (SAEs), or any other safety concerns. No adverse events (AEs) were observed in the 1 and 3 mg/kg dose cohorts. Headache was the most commonly reported treatment-emergent adverse event (TEAE), occurring in 8 of 11 subjects treated with 10 or 30 mg/kg SYNT001. One headache in the 10 mg/kg cohort was moderate (Grade 2) in severity; all other headaches were mild (Grade 1). One mild headache was treated with a single dose of acetaminophen; all other headaches resolved without treatment. Therefore, it is anticipated that the doses selected for this study should be well tolerated and have clinically relevant PD effects in patients with pemphigus.

Further consideration was given to the desired level of FcRn blockade to achieve suppression of IgG to a range that has been previously correlated with disease remission induced by immunoadsorption in autoimmune disorders such as pemphigus vulgaris and myasthenia gravis (ie, >50% decrease in total IgG from baseline) (Blaha et al., 2011; Eming and Hertl, 2006; Kohler et al., 2011).

The Sponsor also considered the potential effects of inhibiting FcRn function as they relate to IC associated innate and adaptive immunity. From the NHP studies, single doses of SYNT001 produced a dose-dependent decrease in total IgG and a further decrease was seen with repeated weekly doses up to a maximum of 70% reduction at 100 mg/kg. This magnitude of total IgG reduction is approaching the expected maximal 90% inhibition of FcRn function based on murine studies performed by the Sponsor and others (Nixon et al., 2015; Roopenian et al., 2003). In the recently completed Phase 1a trial with SYNT001 in healthy volunteers a single dose caused a maximum average 50% drop in total IgG with IV dosing at 30 mg/kg. Based on the

 Syntimmune, Inc.

NHP studies further reductions are expected following multiple dosing. A corresponding decrease in pathogenic autoantibodies is anticipated.

A semi-mechanistic model of FcRn-IgG interactions and FcRn inhibition with SYNT001 was jointly developed by Applied BioMath and the Sponsor. The model was designed to simulate PK and PD responses to various dosing regimens of SYNT001 to inform clinical trial design. Initial simulations were able to capture both PK and PD responses to single doses of SYNT001 from a single-ascending dose study in healthy volunteers and predict multiple dose responses from ongoing studies with good fidelity. The model predicted an IgG reduction of approximately 75% by Day 33, which was determined to be acceptably close to the actual mean IgG reduction of 59% by Day 30 observed in patients. Subsequent iterations of the model have used patient data from ongoing patient studies to further calibrate dose responses. In the most recent simulations, multiple dosing scenarios have been explored, including responses to weekly, bi-weekly, and loading doses. A simulated dosing regimen consisting of three weekly loading doses of 30 mg/kg SYNT001 followed by every other week maintenance doses of 10 mg/kg SYNT001 achieved a nadir IgG reduction of approximately 78% between Days 21 and 28 and maintained an IgG reduction between approximately 50% and 68%. This level of total IgG reduction has been associated with clinical efficacy in early studies of SYNT001-treated pemphigus subjects, and represents a target for future studies in other indications. This regimen of 30 mg/kg loading doses and 10 mg/kg maintenance doses was determined to be the optimal starting regimen to achieve meaningful IgG reduction while maximizing patient safety. Future cohorts may increase the maintenance doses to 20 mg/kg SYNT001, which the model predicts will achieve greater IgG reductions between approximately 55% and 72%. Given the rigorous biological approach taken in the development of the model, simulations of dosing schedules can be considered reliable for the purpose of planning clinical trials.

Several recently completed non-clinical studies support the proposed Cohort 2 dose and dosing regimen. A recently completed 27-week dose-response good laboratory practice (GLP) toxicology study in non-human primates assessed the long-term safety, toxicology, and toxicokinetics of weekly doses of SYNT001. Twenty-seven (27) once weekly 10-minute infusions of SYNT001, at doses of 5, 30, or 100 mg/kg, to cynomolgus monkeys was associated with non-adverse test article-related clinical effects and clinical pathology observations at ≥5 mg/kg. SYNT001 produced dose-dependent reduction of serum IgG levels without affecting IgA, IgM or albumin levels. The NOAEL of SYNT001 was 100 mg/kg following 17 infusions and 30 mg/kg following 27 infusions.

As indicated above, in the recently completed Phase 1a healthy male volunteer study, single doses of SYNT001 up to and including 30 mg/kg have been well tolerated. There were no dose limiting toxicities (DLTs), serious adverse events (SAEs), or any other safety concerns identified. No adverse events (AEs) were observed in the 1 and 3 mg/kg dose cohorts. The only moderate (Grade 2) AE observed was a single instance of headache in the 10 mg/kg cohort. Other subjects had mild (Grade 1) AEs at 10 mg/kg. In Cohort 4 (30 mg/kg), five subjects received SYNT001. All five subjects experienced AEs; all were mild (Grade 1), transient and resolved spontaneously without intervention. The most commonly reported AEs were headache.

A preliminary assessment of safety was conducted by SYNT001 Pemphigus Study SYNT001-103 Dose Escalation Committee (DEC). Seven subjects with pemphigus were treated with

10 mg/kg IV weekly doses over a period of 5 weeks. Overall, SYNT001 10 mg/kg IV was well tolerated. Headache (Grade 1 or 2, self-limited) was the only drug-related AE that was reported in more than one subject. Total IgG and CIC biomarkers were reduced by 59% and 50% respectively, from baseline levels following the fifth dose, returning to baseline within 1 to 2 months. Additionally, preliminary evidence of clinical efficacy as measured by a clinically validated scoring metric, the Pemphigus Disease Area Index, was observed across the population. The DEC approved a dose escalation of SYNT001 from 10 mg/kg IV weekly doses for 5 weeks to 30 mg/kg IV weekly doses for 5 weeks.

Given these preliminary data in non-clinical toxicology species and human subjects, as well as supporting evidence from the computational model, it is anticipated that the doses and dose regimens selected for this study will be well tolerated and will demonstrate clinically relevant pharmacodynamic effects and efficacy in patients with pemphigus. For a summary of findings from the single dose clinical study in healthy subjects and further details regarding the nonclinical findings, please refer to the SYNT001 Investigators Brochure.

## 2.3 Compliance Statement

This study will be conducted in compliance with Good Clinical Practice (GCP), including the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Guidelines and Food and Drug Administration (FDA) regulations, consistent with the principles outlined in the Declaration of Helsinki. In addition, the Investigator agrees to adhere to all applicable local laws and regulatory requirements relevant to the use of new therapeutic agents.

The study will be conducted in compliance with the protocol. The appropriate Institutional Review Boards (IRBs) must approve the protocol, any amendments, and the subject informed consent form (ICF) prior to implementation.

Freely given written informed consent must be obtained from every subject prior to participation in this clinical trial. As part of this procedure, the Investigator must explain orally and in writing the nature, duration, and purpose of the study, and the action of the drug in such a manner that the study subject is aware of the potential risks, inconveniences, or AEs that may occur. The study subject should be informed that he/she is free to withdraw from the study at any time. He/she will receive all information that is required by federal regulations and ICH guidelines. The Investigator or designee will provide the Sponsor with a copy of the IRB-approved informed consent form prior to the start of the study. The rights, safety, and well-being of participating subjects are the most important considerations and should prevail over interests of science and society.

Study personnel involved in conducting this trial will be qualified by education, training, and experience to perform their respective task(s). This trial will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

# 3. STUDY OBJECTIVES AND ENDPOINTS

| Primary Objectives | Primary Endpoints |
|---|---|
| Safety: To evaluate the safety of IV infusions of SYNT001 at different dose levels and dosing regimens in subjects with pemphigus (vulgaris or foliaceus) | Safety: The evaluation of SYNT001 safety based on vital signs, physical examinations, electrocardiograms (ECGs), clinical safety laboratory tests, the incidence of adverse events (AEs), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) summarized by dose and dosing regimen, severity, and relationship to study drug |
| Dose Selection: To determine a MED of SYNT001 as assessed by (i) total IgG level nadir and (ii) the proportion of subjects that meet the criteria for response by Pemphigus Disease Area Index total activity score (PDAI) | Dose Selection: The determination of dose and dosing regimen of SYNT001 that achieves (i) total IgG level nadir decrease by ≥60% and ≤90% from baseline and (ii) a PDAI total activity score of ≥50% reduction from baseline to allow further clinical development in subjects with pemphigus (vulgaris or foliaceus) |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the efficacy of doses of SYNT001 at different dose levels and dosing regimens on pharmacodynamics (PD) biomarkers | The evaluation of PD biomarkers based on absolute serum levels and percent change from baseline of total IgG, IgG subtypes (IgG1-4), immunoglobulin A (IgA), immunoglobulin M (IgM), albumin, and CIC summarized by dose, dosing regimen and visit |
| To determine the pharmacokinetics (PK) of SYNT001 following IV infusions at different dose levels and dosing regimens | The determination of PK parameters including half-life ( $t_{1/2}$ ), maximum serum concentration determined directly from the concentration-time profile ( $C_{max}$ ), observed time of peak serum concentration ( $T_{max}$ ), area under the serum concentration-time curve from pre-dose (time <sub>0</sub> ) to 24 hours post-dose (AUC <sub>0-24</sub> ), and area under the serum concentration-time curve from pre-dose (time <sub>0</sub> ) to infinity (AUC <sub>0-<math>\infty</math></sub> ), (Cohort 1); maximum serum concentration determined directly from the maximum serum concentration and corresponding $T_{max}$ (Cohort 2 onwards) summarized by dose, dosing regimen, visit and time point |
| To assess the efficacy of doses of SYNT001 at different dose levels and dosing regimens on disease markers | <ul> <li>The assessment of pemphigus disease activity by responses on the PDAI based on absolute and percent change from baseline, summarized by dose, dosing regimen and visit</li> <li>The assessment of pemphigus disease activity by pathogenic antibody levels based on absolute and percent change from baseline of serum anti-desmoglein 1 and 3 antibody (anti-Dsg 1 and anti-Dsg</li> </ul> |

| | 3) levels summarized by dose, dosing regimen and visit |
|---|---|
| To measure the immunogenicity of SYNT001 administered at different dose levels and dosing regimens | The immunogenicity of SYNT001 as determined by presence of anti-SYNT001 binding antibodies and neutralizing antibodies summarized by dose, dosing regimen, visit and time point |
| <b>Exploratory Objectives</b> | <b>Exploratory Endpoints</b> |
| To explore the effect of SYNT001 at different dose levels and dosing regimens on biomarkers to understand the pathophysiology of the disease and the SYNT001 mechanisms of action | The exploration of SYNT001 mechanisms of action and effects of SYNT001 on pathophysiology summarized by dose, dosing regimen and visit as determined by: |
| | <ul> <li>Complement component 3 levels by nephelometry</li> <li>Anti-epithelial cell antibody (AECA) titers by indirect immunofluorescence</li> <li>Fc gamma R2A receptor (FCGR2A) single nucleotide polymorphisms (SNP) by genotyping</li> <li>Presence of disease and inflammatory markers by total RNA sequencing</li> <li>Immunophenotyping including measurements of T cells, monocytes, natural killer (NK) cells and B cells by flow cytometry</li> <li>Urine IgG levels to explore SYNT001 distribution and elimination (Cohort 1 only)</li> <li>Exploratory biomarkers to investigate immune response associated with pemphigus</li> </ul> |
| To determine the impact of different SYNT001 dose levels and dosing regimens on the subject's use of corticosteroids to treat their pemphigus (vulgaris or foliaceus) | The evaluation of corticosteroid use during the study will be summarized by dose, dosing regimen and visit |
| To assess the impact of SYNT001 on the subject's health-related quality of life (HR-QoL) at different dose levels and dosing regimens | The assessment of SYNT001 impact on subject's health-related quality of life (HR-QoL) by responses to the Autoimmune Bullous Diseases Quality of Life (ABQoL) questionnaire and Skindex-29 scores summarized by dose, dosing regimen and visit |
| To assess the effect of SYNT001 on the appearance of skin and mucosal lesions at different dose levels and dosing regimens | The qualitative assessment of changes in appearance of skin and mucosal lesions as determined by photography presented by dose, dosing regimen and visit |
| To quantify the amount of SYNT001 in skin (skin biopsies optional) | The determination of SYNT001 levels in skin biopsies across timepoints (skin biopsies optional) (Cohort 1 only) |

#### 4. STUDY DRUG

#### 4.1 Description of SYNT001

SYNT001 is provided in vials containing 5 mL SYNT001 (extractable volume) at a nominal concentration of 50 mg/mL. The product is supplied as a liquid at pH  $6.5 \pm 0.5$ . SYNT001 is diluted in dextrose 5% in water (D5W) to prepare the solution for infusion. SYNT001 will be infused via IV in 250 mL over 1 hour  $\pm$  15 minutes using a 0.2-micron, inline filter.

Investigators may adjust the duration of the infusion if needed to improve tolerability. Infusion of SYNT001 should be completed within 4 hours of preparation as described in the Pharmacy Manual. For detailed information regarding SYNT001 preparation and administration, refer to the Pharmacy Manual.

#### 4.2 Dose Requirements

The specification for host cell deoxyribonucleic acid (DNA) in SYNT001 is <2 pg/mg, the limit of quantitation of the assay. To comply with regulatory guidelines, which specify a maximum level of 10 ng host cell DNA per dose, dosing per subject is limited to 5000 mg SYNT001.

For example, a subject with a body weight of 166 kg and enrolled in the ≤30 mg/kg dose cohort will receive ≤4960 mg SYNT001 per dose. If a subject's body weight extrapolates to an expected dose ≥5000 mg SYNT001, the dose will be capped at 5000 mg to ensure the 5000 mg SYNT001 per dose limit is not exceeded.

#### 4.3 Handling and Storage of SYNT001

All supplies of SYNT001 will be provided by the Sponsor and must be stored refrigerated (2°C to 8°C/36°F to 46°F) in the carton and protected from light, in a securely locked area, accessible to authorized persons only, until needed for dose preparation.

### 4.4 Study Drug Accountability

The Investigator (or designee) is responsible for maintaining accurate accountability records of the study drug throughout the clinical study. Qualified site personnel will inventory the study drug received and will maintain records of disposition of the drug, including dates, quantity and use. All study drug received at the site must be accounted for on an accountability log provided by the Sponsor. All dispensing and accountability records will be available for Sponsor review. Study drug accountability will be verified during on-site monitoring visits.

Upon the completion or termination of the study, and upon written authorization from the Sponsor, or its representative, all unused and/or partially used study drug should be returned or destroyed at the investigational site, as specified by Sponsor. It is the Investigator's responsibility to ensure that the Sponsor, or its representative, has provided written authorization that procedures for proper disposal of the study drug have been established, and that appropriate records of the disposal are documented and maintained. No unused study drug may be disposed of until fully accounted for by the Sponsor monitor (or designee).

#### 5. STUDY DESIGN

#### 5.1 Study Sites

This study will be conducted at approximately 20 global study sites.

#### 5.2 Overview of Study Design

This is a multicenter, open-label safety study to determine the dose regimen of SYNT001 administered IV in subjects with pemphigus (vulgaris or foliaceus). Up to 8 subjects with a diagnosis of pemphigus (vularis or foliaceus) will receive SYNT001 10 mg/kg weekly x 5 doses (Cohort 1).

Up to 12 subjects with a diagnosis of pemphigus (vulgaris or foliaceus) will receive SYNT001 30 mg/kg weekly x 3 doses (Loading), followed by SYNT001 10 mg/kg every other week x 5 doses (Maintenance) (Cohort 2) (Figure 1). Subjects in each cohort will complete the following periods of assessment: Screening, Treatment, and Follow-Up.

For Cohort 1 details of the dosing schedule and assessments, see Table 2. For Cohort 2 details, see Table 3.

The Dose Escalation Committee (DEC) will consist of the Medical Monitor, an Independent Clinical Expert and the Sponsor Medical Lead. The DEC may request that Investigators, other experts, or members within their organization participate in the review. Additional information on the DEC's responsibilities is provided in Section 9.5 and the DEC Charter.

An overview of the study cohorts is provided in Table 4 and Figure 1 shows a schematic of the study design.

| Cohort No. | No. of Subjects | SYNT001 Dose | No. of Doses | Frequency of Doses |
|---|---|---|---|---|
| 1 <sup>a</sup> | Up to 8 | 10 mg/kg | 5 | Weekly |
| 2 <sup>b</sup> | Up to 12 | Loading:<br>30 mg/kg <sup>c</sup> | 3° | Weekly <sup>c</sup> |
| | | Maintenance:<br>10 mg/kg <sup>c</sup> | 5° | Every other week <sup>c, d</sup> |

Table 4. Cohort Overview

- a. No more than 3 subjects with pemphigus foliaceus may be enrolled
- b. Two or fewer subjects with pemphigus foliaceus may be enrolled
- c. The dose, number of doses, and frequency of doses in Cohort 2 will be confirmed based on review of safety and PD evaluations, including but not limited to, dose-limiting toxicities, AEs, TEAEs, SAEs, and total IgG levels. Following Sponsor review of emerging safety, PD and efficacy data, the Loading dose may be reduced to 20 or 10 mg/kg weekly and/or the Maintenance dose may be increased to 20 or 30 mg/kg every other week and/or dose frequency may be increased to weekly.
- d. Ongoing safety and PD evaluations may result in modification of the dose and dosing regimen in Cohort 2. See APPENDIX 5 for the corresponding visit schedule.
Subjects will be enrolled at staggered intervals to facilitate adequate safety evaluation before dosing of subsequent subjects

At 24-hour and 7-day intervals described below, all available safety data (including but not limited to dose-limiting toxicities [DLTs], AEs, TEAEs, SAEs, and PD (including but not limited to IgG levels), will be reviewed.

### Safety Review of 24-hour Data

The first 2 subjects in each cohort will be dosed at least 24 hours apart. A DEC review of the 24-hour safety data for the first subject in Cohort 1 will be performed to ensure that there are no overt safety concerns before dosing the second subject. The Sponsor Medical Lead and Medical Monitor will conduct the 24-hour safety data review for the first subject in Cohort 2.

### Safety Review of 7-day Data

The 7-day safety data for the first 2 subjects in Cohort 1 will be reviewed by the DEC prior to dosing the remaining subjects in the cohort. The Sponsor Medical Lead and Medical Monitor will conduct the 7-day safety data review in Cohort 2.

The 24-hour and 7-day reviews will consider seriousness and severity of AEs/TEAEs/SAEs and relatedness to study drug, vital sign assessments, physical examinations, and clinical laboratory testing.

For further information about dose escalation and study stopping rules, refer to Section 9.5.1 and Section 9.5.2, respectively.

### 5.3 Randomization and Blinding

This is an open-label study.

## 5.4 Duration of Subject Participation

The duration of subject participation for each cohort is as follows:

| Cohort | Screening | Treatment | Follow-up | Maximum Total | |
|--------|-----------|-----------|-----------|---------------|----------|
| | | | | Days | Weeks |
| 1 | ≤14 days | 28 days | 84 days | 126 days | 18 weeks |
| 2 | ≤14 days | 84 days | 56 days | 154 days | 22 weeks |

### 6. STUDY POPULATION

## 6.1 Target Population

This study will be conducted in male and female subjects aged 18 and older with a confirmed diagnosis of pemphigus (vulgaris or foliaceus). Subjects will be enrolled only once in the study and will not be included in subsequent dosing cohorts. Subjects who withdraw for any reason other than an AE may be replaced.

Within Cohort 1, no more than 3 subjects may be enrolled with pemphigus foliaceus. Within Cohort  $2, \le 2$  subjects with pemphigus foliaceus may be enrolled.

### 6.2 Inclusion Criteria

A subject must meet the following criteria to be eligible for the study:

- 1. Willing and able to read, understand, and sign an informed consent form.
- 2. Male or female  $\geq$ 18 years of age at the time of screening.
- 3. Documented diagnosis of pemphigus vulgaris or foliaceus based on all 3 of the following criteria:
  - a. Documented clinical history consistent with pemphigus vulgaris or foliaceus (clinical presentation defined as mucosal and/or skin lesions).
  - b. Presence of Anti-Dsg 1 or 3 antibodies above the upper limit of normal (ULN).
  - c. History of at least one positive tissue-based test (eg, biopsy, direct immunofluorescence [DIF]).
- 4. Active disease defined as lesions lasting >2 weeks, and 3 active lesions in skin or mucosa or 2 active lesions with at least one being a skin lesion >1 cm diameter:
  - a. If treated with rituximab or other anti-CD20 mAb, last dose >9 months prior to screening.
  - b. If being treated with other immunosuppressants (ie, azathioprine, mycophenolate mofetil, methotrexate, dapsone, cyclosporine, tacrolimus, sirolimus, or low-dose cyclophosphamide [ $\leq$ 100 mg/day]), dose must be stable, defined as  $\leq$ 25% change in dose, for 4 weeks prior to screening.
  - c. On stable dose of corticosteroids, defined as  $\leq 1$  mg/kg of prednisone or equivalent and may not be increased by more than 50% in the 2 weeks prior to screening.
  - d. Allowed topical therapies for pemphigus lesions upon entering the study include petroleum jelly or Aquaphor® for the skin or chlorhexidine for the mouth.
  - e. Stable use of topical low strength hydrocortisone (≤1%), tacrolimus, sirolimus, or pimecrolimus for lesions contributing <10% of the PDAI total activity score for the 4 weeks prior to screening is allowed. Stable use of dexamethasone elixir solution (swish and spit only) for oral lesions for the 4 weeks prior to screening is allowed.
  - f. If not on regular corticosteroids, no pulse corticosteroids are allowed in the 2 weeks prior to screening.
- 5. Body mass index (BMI)  $> 18.5 \text{ kg/m}^2$ .
- 6. Has a negative pregnancy test documented prior to the first dose of study drug (for women of childbearing potential).

- 7. Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception (<1% per year failure rate) from the screening period through the final study visit: oral contraceptive, condom with or without spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or intrauterine device (IUD). A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception.
- 8. Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months do not require contraception during the study.
- 9. Males with female partners of childbearing potential, including males who are surgically sterile (post vasectomy), must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through the final study visit.
- 10. A PDAI total activity score of >4 at screening.

### 6.3 Exclusion Criteria

A subject who meets any of the following criteria is ineligible for the study:

- 1. Subject unable or unwilling to comply with the protocol.
- 2. Active non-hematologic malignancy or history of non-hematologic malignancy in the 3 years prior to screening (exclusive of non-melanoma skin cancer and cervical cancer in situ).
- 3. Positive for human immunodeficiency virus (HIV) or hepatitis C antibody.
- 4. Positive for hepatitis B surface antigen.
- 5. Active infection or history of recurrent infections.
- 6. IVIG treatment within 30 days of screening.
- 7. Received any cytotoxic (other than azathioprine) or any non-anti-CD20 mAb therapy in the 3 months prior to screening.
- 8. Any exposure to an investigational drug or device within the 30 days prior to screening.
- 9. Plasmapheresis or immunoadsorption within 30 days of screening.
- 10. Cellular therapy, including chimeric antigen receptor and T-cell (CAR-T), at any time prior to screening.
- 11. Use of any systemic or topical immunosuppressive drugs within 3 months of screening not including dose allowed by the inclusion criteria.
- 12. Serum total IgG <600 mg/dL at screening.
- 13. Subject has any current medical condition that, in the opinion of the Investigator, may compromise their safety or compliance, preclude successful conduct of the study, or interfere with interpretation of the results (eg, a significant pre-existing illness or other major comorbidity that the Investigator considers may confound the interpretation of the study results).
- 14. Any vaccination within 2 weeks of screening.

### 7. STUDY PROCEDURES

### 7.1 Informed Consent

All subjects must take part in the informed consent process. Adequate time must be allowed for the subject to ask questions and make a voluntary decision. No protocol-specific procedures, including screening procedures are to be performed until the subject has signed and dated an IRB-approved ICF. Subjects may withdraw consent at any time. Participation in the study may be terminated at any time without the subject's consent as determined by the Investigator.

## 7.2 Demographics and Medical History

Demographics (age, gender, race and ethnicity) and medical history will be obtained from the subject and recorded on the source document and electronic case report form (eCRF). Medical history will capture the subject's current medical history (current disease processes), past medical status (past disease processes), history of surgery, concomitant treatments, and relevant clinical response to past disease specific treatments including duration and dosing of such treatments.

## 7.3 Physical Examination

A complete physical examination will include measurements of weight (in kg) and height (in cm; height to be measured only at screening visit) and a review of the following body systems:

- General appearance
- Head, eyes, ears, nose, and throat
- Neck
- Respiratory
- Cardiovascular
- Abdomen
- Neurologic
- Extremities
- Dermatologic
- Lymphatic

Any abnormal and clinically significant findings from the physical examination must be recorded in the appropriate eCRF. Findings at screening and Day 0 (pre-dose) will be recorded as medical history.

## 7.4 Vital Sign Measurements

Vital sign assessments will include measurements of sitting blood pressure (mm Hg), heart rate (beats per minute), respiration rate (breaths per minute), pulse oximetry, and oral temperature (Celsius). Abnormal results are to be repeated after 5 minutes of rest. See Table 5 for timing window allowances with respect to measurement collection.

When vital signs are to be collected at the same time point as a blood collection, vital signs should be collected first. Vital sign measurements will be collected after the subject has been sitting for 5 minutes. Subjects should be seated quietly for at least 5 minutes in a chair with their backs supported, their feet flat on the floor (legs uncrossed), and their arms bared on a hard surface, with the arm slightly abducted and bent, with palm up and the midpoint of upper arm at heart level. Correct cuff and bladder size should be utilized and the same cuff and arm should be used per subject throughout study.

Vital sign measurements are to be obtained immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; 30 minutes, 1 hour, and 2 hours following completion of the infusion. Abnormalities in vital sign measurements will be graded in severity per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) scale Version 4.03.

Table 5. Timing window allowances for PK/PD sampling, ECG, and vital sign measurements at dosing visits

| Time Point | Tolerance Window | |
|---|---|---|
| | Cohort 1 | Cohort 2 |
| Pharmacokinetic Sampling | | |
| 0 hour | -240 minutes to 0 hour | -240 minutes to 0 hour |
| 5 minutes post end-of-infusion | ±5 minutes | ±5 minutes |
| 1 hour post end-of-infusion | N/A | ±15 minutes |
| 2 hours post end-of-infusion | $\pm 15$ minutes | ±15 minutes |
| 4 and 6 hours post end-of-infusion | $\pm 15$ minutes | N/A |
| 24 hours (1 day) post end-of-infusion | ±60 minutes | N/A |
| 48 hours (2 days) post end-of-infusion | ±120 minutes | N/A |
| Pharmacodynamic Sampling | | |
| 0 hour | -240 minutes to 0 hour | -240 minutes to 0 hour |
| 24 hours (1 day) post end-of-infusion | ±60 minutes | N/A |
| 48 hours (2 days) post end-of-infusion | ±120 minutes | N/A |
| ECG | | |
| 5 minutes post end-of-infusion | ±10 minutes | ±10 minutes |
| Vital Signs <sup>a</sup> | | |
| 0 hour | -240 minutes to 0 hour | -240 minutes to 0 hour |
| 15, 30, and 45 minutes after start of infusion | ±5 minutes | ±5 minutes |
| At completion of the infusion | ±10 minutes | ±10 minutes |
| 30 minutes, 1 and 2 hours post end-of-infusion | ±10 minutes | ±10 minutes |

## 7.5 Clinical Laboratory Measurements

Laboratory testing (hematology, urinalysis, serum chemistry, virology, serology, pregnancy tests, PD, PK, and ADAs) will be performed using established methods by a central laboratory. Clinical safety laboratory panels are listed in Table 6. Blood and urine for hematology, serum chemistry, and urinalysis will be prepared using standard procedures. Results will be provided to the Investigator. Aliquots from the PK, biomarker and ADA samples may be retained as back-up for additional testing as necessary. Subjects will be in a seated or supine position during blood collection. Collection times for all safety, PD, and exploratory labs are outlined in Table 2 and Table 3.

Table 6. Clinical Safety Laboratory Panels

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| <ul> <li>CBC with differential and blood smear</li> <li>Erythrocyte sedimentation rate</li> </ul> | <ul> <li>Albumin</li> <li>Alkaline phosphatase</li> <li>ALT</li> <li>AST</li> <li>BUN</li> <li>C-Reactive Protein</li> <li>Calcium</li> <li>Carbon dioxide</li> <li>Chloride</li> <li>Creatinine</li> <li>Glucose</li> <li>LDH</li> <li>Phosphorus</li> <li>Potassium</li> <li>Sodium</li> <li>Total and direct bilirubin</li> <li>Total protein</li> <li>Uric acid</li> </ul> | <ul> <li>Appearance</li> <li>Color</li> <li>pH</li> <li>Specific gravity</li> <li>Ketones</li> <li>Protein</li> <li>Glucose</li> <li>Nitrite</li> <li>Urobilinogen</li> <li>Blood/hemoglobin</li> <li>Leukocyte esterase</li> <li>Bilirubin</li> <li>Microscopic examination of sediment: only if the results of the urinalysis dipstick evaluation are positive for blood/hemoglobin</li> </ul> |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; CBC = complete blood count; HIV = human immunodeficiency virus; LDH = lactate dehydrogenase; VZV = Varicella-Zoster virus.

Abnormalities in clinical laboratory tests that are considered clinically significant are to be recorded on the AE eCRF page. Laboratory results will be graded using the NCI CTCAE, Version 4.03. If laboratory values constitute part of an event that meets criteria defining it as serious, the event (and associated laboratory values) must be reported as an SAE (see Section 10.2.3).

### 7.5.1 Pregnancy Testing

Pregnancy testing will be performed for women of childbearing potential. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.

## 7.5.2 Virology

Testing for hepatitis C antibody, hepatitis B surface antigen, and HIV antibody will be performed at screening.

## 7.5.3 Serum Tetanus Antibody and Varicella-Zoster Virus Antibody Testing

Samples for serum tetanus antibody and VZV antibody testing are to be collected. Any subject whose baseline value for tetanus or VZV was above the protective level at baseline, and is not within 30% of the baseline value or is below the protective level by the end-of-study visit, will be referred to their primary care physician for further management.

### 7.5.4 Pharmacokinetics (PK) Sampling

The following PK parameters will be studied in Cohort 1:  $t_{1/2}$ ,  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-24}$ , and  $AUC_{0-\infty}$ . For Cohort 2, the PK parameters studied will be  $C_{max}$  and  $T_{max}$ . For Cohort 2, the PK parameters studied will be maximum serum concentration of SYNT001 and the associated  $T_{max}$ .

Specific collection times and timing window allowances are detailed in Table 5. Detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

## 7.5.5 Pharmacodynamic Sampling

PD samples will be collected for analyses throughout the study. Measurements for albumin will be derived from the clinical safety laboratory results. Specific collection times are detailed in. Samples for each type of PD will be collected according to the schedule shown in Table 7.

Table 7. Pharmacodynamic Assessments

| Parameter | <b>Collection Time Points</b> | |
|---|---|---|
| | Cohort 1 | Cohort 2 <sup>a</sup> |
| Immunoglobulins: • IgG • IgG subtypes (IgG1-4) • IgA • IgM | Screening and Days 0, 1, 2, 5, 7, 12, 14, 19, 21, 28, 29, 30, 33, 42, 56, 84, and 112 | Screening and Days 0, 7, 14, 28, 42, 56, 70, 84, 91, 112, and 140 |
| Circulating immune complexes (CIC) | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84, and 112 | Days 0, 7, 14, 28, 42, 56, 70, 84, 91, 112, and 140 |
| Albumin | Screening and Days 0, 7, 14, 21, 28, 33, 42, 56, 84, and 112 | Screening and Days 0, 7, 14, 28, 42, 56, 70, 84, 91, 112 and 140 |
| Anti-Dsg (1 and 3) antibody<br>titers | Screening and Days 0, 7, 14, 33, 56, 84, and 112 | Screening and Days 0, 7, 14, 28, 42, 56, 70, 84, 91, 112, and 140 |
| C3 and AECA levels by<br>indirect immunofluorescence | Days 0, 14, 33, 56, 84, and 112 | Screening and Days 0, 7, 14, 28, 42, 56, 70, 84, 91, 112, and 140 |
| Exploratory biomarkers (RNAseq, urine IgG) <sup>b</sup> | Days 0, 14, 33, 56, 84, and 112 | Days 0, 28, and 91 |
| Immunophenotyping by flow<br>cytometry for measurement of<br>T cells, monocytes, NK cells,<br>and B cells | Days 0, 28, and 56 | Days 0, 28, and 91 |
| Exploratory biomarker (FCGR2A SNP, via buccal swab) | Day 0 | Day 0 |
| Exploratory pemphigus<br>immune response biomarkers | Days 0, 5, 7, 12, 14, 19, 21, 28, 33, 42, 56, 84, and 112 | Days 0, 7, 14, 28, 42, 56, 70, 84, 91, 112, and 140 |

<sup>&</sup>lt;sup>a</sup> Ongoing safety and PD evaluations may result in modification of the dosing regimen from every other week to weekly. See APPENDIX 5 for the corresponding visit schedule.

See Table 5 for timing window allowances with respect to measurement collection. More information, including detailed instructions for sample collection (including collection tubes) and preparation will be provided in a separate laboratory manual.

### 7.5.6 Immunogenicity Testing

SYNT001 is being developed for the acute and chronic therapy of autoimmune disorders. Although SYNT001 is a humanized IgG4 mAb, exposure to SYNT001 in clinical trials could result in the development of ADAs, with potential consequences ranging from neutralization with possible lessening of drug efficacy to safety consequences such as allergic reactions. Testing will first detect binding ADAs. Then, for all confirmed positive samples, an ADA titer will be determined and there will be testing for neutralizing antibodies using a validated cell-based assay.

More information, including detailed instructions for sample collection and preparation will be provided in a separate laboratory manual.

<sup>&</sup>lt;sup>b</sup> Urine IgG collected in Cohort 1 only.

## 7.6 12-Lead Electrocardiogram (ECG)

On dose administration days, digital 12-lead ECG measurements will be obtained at 5 minutes after the completion of the infusion. When ECGs are to be collected at the same time point as a blood collection, ECGs should be collected first. All ECGs are to be performed with the subject in a supine position having rested in this position for at least 5 minutes before each reading. ECGs are to be performed in triplicate, each at an interval of 1 to 2 minutes apart (Cohort 1) or approximately 1 minute apart (Cohort 2). See Table 5 for timing window allowances with respect to performing ECG.

The following ECG parameters will be collected: PR interval, RR interval, QRS interval, and QT interval. The ECG findings will be evaluated by a qualified physician for the presence of abnormalities (qualitative assessment). The physician will assess each ECG as normal, abnormal/not clinically significant, or abnormal/clinically significant.

Normal corrected QT interval using Fridericia's formula (QTcF) is ≤450 msec.

Abnormalities in the ECG that appear following therapy or that result in clinical signs and symptoms are considered clinically significant for the purposes of this study and will be recorded on the AE eCRF.

## 7.7 Pemphigus Disease Area Index (PDAI)

Pemphigus severity and disease activity will be measured using the PDAI in regions where a validated questionnaire is available. A PDAI total activity score will be determined at screening. To be eligible for study participation, the patient's grade by disease severity must be >4. Assuming subject eligibility, the PDAI will be administered during Treatment Period and Follow-up Period. Disease severity categories by PDAI are mild (0 to 8), moderate (9 to 24), and severe ( $\geq$ 25) (Shimizu et al., 2014). The Investigator will determine a PDAI score as follows: 0 to 250 points for disease activity ( $\leq$ 120 for skin,  $\leq$ 10 for scalp, and  $\leq$ 120 for mucosa), and 0 to 13 points for damage ( $\leq$ 12 for skin and  $\leq$ 1 for scalp) (Rosenbach et al., 2009). See Appendix 2.

### 7.8 Study Drug Administration

SYNT001 will be given as a 250-mL IV infusion over 1 hour  $\pm$  15 minutes using a 0.2-micron, inline filter.

## 7.9 Photographs

Photographs will be taken of active lesions and follow-up photographs will be taken of the same areas at timepoints indicated in Table 2 and Table 3. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made. A separate manual describing the procedures for taking photographs will be provided.

### 7.10 Health-Related Quality of Life Assessments

For Cohort 2, health-related quality of life will be assessed using ABQoL and Skindex-29 in regions where a validated questionnaire is available. The ABQoL questionnaire was developed

 Syntimmune, Inc.

in Australia as a patient-based measure to quantify disease burden, monitor disease activity and evaluate response to therapeutic intervention in patients with autoimmune bullous disease (Sebaratnam et al., 2013; Sebaratnam et al., 2015) (Appendix 3). Skindex-29 was developed to measure the effects of skin disease on patients' quality of life using a self-administered 30-question dermatology survey (Chren et al., 1996) (Appendix 4).

### 7.11 Adverse Event Assessments

Information regarding the occurrence of AEs will be collected from the time the subject signs the informed consent form and continuing through the last study visit. Findings at screening and Day 0 (pre-dose) will be recorded as medical history. Any known untoward event that occurs beyond the AE reporting period that the Investigator assesses as related to study drug also should be reported as an AE. Clinical AEs will be graded using the NCI CTCAE, Version 4.03 (Appendix 1).

**Note:** AEs resulting in a subject's permanent discontinuation from the study, regardless of seriousness or relationship to study drug, MUST be promptly reported to the Sponsor. Additionally, subjects must be followed until return to normal and/or resolution of the AE.

See Section 10 for more information.

### 7.12 Prior and Concomitant Medications

All treatments a subject receives within 14 days prior to enrollment through the end of the study will be documented on the source document and eCRF. A history of treatments taken for the primary disease, even if not taken within the 14 days prior to enrollment, will be collected.

### **Permitted Medications**

Concomitant medication and treatment for co-existing conditions, including those for pemphigus, are permitted if not listed as prohibited.

- 1. Topical antibiotics to treat active infections that occur during the study.
- 2. Topical or systemic treatments for oral candidiasis.
- 3. Topical lidocaine for transient pain relief as needed.
- 4. Concomitant treatment that is medically indicated for any AEs the subject experiences during the study.
- 5. Medication for potential infusion-related reactions (IRRs) including post-infusion headache: The Investigator may recommend prophylactic use of acetaminophen, IV hydration, diphenhydramine, histamine<sub>2</sub> (H<sub>2</sub>) blockers (eg, ranitidine, famotidine), etc to manage potential IRRs.
- 6. Low-strength corticosteroids (eg, hydrocortisone ≤1%) applied to a single lesion contributing <10% of the PDAI total activity score.
- 7. Topical tacrolimus, sirolimus or pimecrolimus applied to a single lesion contributing <10% of the PDAI total activity score.
- 8. Dexamethasone elixir solution for oral lesions if dose remains stable throughout trial participation (swish and spit only).

 Syntimmune, Inc.

9. Stable regimen of the following systemic immunosuppressants: azathioprine, mycophenolate mofetil, methotrexate, dapsone, cyclosporine, tacrolimus, sirolimus, corticosteroids, or low dose oral cyclophosphamide (≤100 mg/day).

Fourteen days after the final dose of SYNT001, corticosteroids may be tapered at the Investigator's discretion.

#### **Prohibited Medications**

Use of the following medications will not be permitted during the study unless specified above as permitted:

- 1. Rituximab or other anti-CD20 antibody
- 2. Monoclonal antibodies other than study drug
- 3. Any topical or systemic immunosuppressive drugs apart from those that are listed as permitted.
- 4. IV corticosteroids prior to infusion (except in subjects who received corticosteroids for treatment of a prior IRR to SYNT001)
- 5. Any investigational drug or device
- 6. Vaccinations within 2 weeks of screening through 28 days following final dose of study drug

### **Corticosteroids**

### Before enrollment

The dose of corticosteroids taken for pemphigus or any other condition prior to screening must be at a dose  $\leq 1$  mg/kg and the dose level must have not increased in dose level by more than 50% in the 2 weeks prior to screening. No pulse dosing of steroids is permitted in the 2 weeks prior to screening.

### From screening until 2 weeks after the last dose of SYNT001

The dose of corticosteroids taken for pemphigus or any other condition should remain stable (<10% change in dose level) from screening until 2 weeks after the last dose of SYNT001. Corticosteroids should neither be started nor discontinued during this period with the exception of subjects who experience an IRR that requires corticosteroids as part of the management of the IRR. Such subjects may receive corticosteroids prophylactically prior to subsequent SYNT001 infusions at the discretion of the Investigator.

### From 2 weeks after the last dose of SYNT001 until end of study participation

At the discretion of the Investigator, but only after at least 2 weeks beyond the last dose of SYNT001, a slow corticosteroid taper may be started as per the following suggested schedule:

• If on >30 mg of prednisone per day, decrease by no more than 10 mg every two weeks until a final dose.

If per the Investigator's judgement, the subject would benefit from a change to the pemphigus treatment beyond the allowed steroid taper, this will be considered on a case-by-case basis in consultation with the Sponsor.

 Syntimmune, Inc.

## 7.13 Skin Biopsy

In Cohort 1, optional skin biopsy samples from lesional or non-lesional skin will be collected to analyze SYNT001 levels.

### 8. STUDY ASSESSMENTS

Study assessments are performed on a weekly basis and will be comprised of the following periods: Screening, Treatment (including Baseline [Day 0]), and Follow-Up (including End-Of Study). For those subjects that complete all periods in Cohort 1, maximum study duration is 126 days. For those subjects that complete all periods in Cohort 2, maximum study duration is 154 days.

Further detail on specific study assessments is provided in Section 7.

## 8.1 All Cohorts: Screening Period and First Treatment (Day 0)

### 8.1.1 All Cohorts: Screening Period (Day -14 to Day -1)

For all cohorts, informed consent must be obtained before any study-specific samples are taken or study-specific tests or evaluations are conducted. The following assessments at the screening visit are to occur within 14 days before dosing. Study eligibility will be based on satisfying all the study inclusion and exclusion criteria (see Section 6).

At the screening visit, information will be collected and subjects will have clinical evaluations as follows:

- Informed consent
- Medical history and demographic data
- Review inclusion and exclusion criteria
- Complete physical examination, including height and weight
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature); abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI (Cohort 2 only)
- Pregnancy test
- Hepatitis and HIV screen
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position)
- Immunogenicity sample collection (*Cohort 2 only*)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - Anti-Dsg1 and Dsg3 antibody titers
  - C3 (*Cohort 2 only*)
  - AECA (Cohort 2 only)
- Concomitant medication assessment
- AE assessment

### 8.1.2 All Cohorts: Enrollment and First Treatment (Day 0)

For all cohorts, study Day 0 is defined as the date the subject is administered their first dose of study drug. On Day 0, subjects will be asked to come to the clinic and the following procedures will be performed prior to the first dose of study drug:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Cohort 2 only)
- Serum tetanus antibody and VZV antibody
- PDAI
- PK baseline sample collection (collected just prior to the start of the study drug infusion)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - FCGR2A SNP via buccal swab
  - RNAseq
  - Urine IgG (Cohort 1 only)
  - Immunophenotyping
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional) (Cohort 1 only)
- Photography
- HR-QoL assessments (ABQoL, Skindex-29) (Cohort 2 only)

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

## After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

 Syntimmune, Inc.

- PK sample collection at 5 minutes. Thereafter at 2, 4, 6 hours (Cohort 1) or 1 and 2 hours (Cohort 2) after the completion of study drug infusion; record collection date and time for each PK sample
- 12-lead ECG (to be obtained in triplicate approximately 5 minutes after the completion of study drug infusion

### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### 8.2 Cohort 1: Day 1 to 84

### 8.2.1 Cohort 1: Follow-up Day 1

On Day 1 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Skin biopsy (optional)
- Concomitant medication assessment
- AE assessment

### 8.2.2 Cohort 1: Follow-up Day 2

On Day 2 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 0), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Skin biopsy (optional)
- Concomitant medication assessment
- AE assessment

### 8.2.3 Cohort 1: Follow-up Day 5

On Day 5 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 0), subjects may return to the clinic or be visited by an at-home nurse, and the following procedures are to be performed:

 Syntimmune, Inc.

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment

## 8.2.4 Cohort 1: Treatment Day 7 (Dose 2)

On Day 7 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - Exploratory pemphigus immune response biomarkers

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### 8.2.5 Cohort 1: Follow-up Day 12

On Day 12 ( $\pm$  6 hours), subjects may return to the clinic or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- If visit performed at the study site: 12-lead ECG to be obtained in triplicate
- Concomitant medication assessment
- AE assessment

### 8.2.6 Cohort 1: Treatment Day 14 (Dose 3)

On Day 14 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

 Syntimmune, Inc.

## After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

## 8.2.7 Cohort 1: Follow-up Day 19

On Day 19 ( $\pm$  6 hours), subjects may return to the clinic or be visited by an at-home nurse, and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment

### 8.2.8 Cohort 1: Treatment Day 21 (Dose 4)

On Day 21 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers

### After the preceding procedures and assessments are completed:

• Study drug administration (record date and time of dose of study drug)

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

## After administration of study drug, the following post treatment procedures and assessments will be performed:

• Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest

### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### 8.2.9 Cohort 1: Treatment Day 28 (Dose 5)

On Day 28 ( $\pm$  6 hours) subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PK sample collection (collected just prior to the start of the study drug infusion)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Immunophenotyping
  - Exploratory pemphigus immune response biomarkers

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

 Syntimmune, Inc.

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest
- PK sample collection at 5 minutes and 2, 4, and 6 hours after the completion of study drug infusion; record collection date and time for each PK sample
- 12-lead ECG (to be obtained in triplicate at 5 minutes after the completion of study drug infusion

### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### **8.2.10** Cohort 1: Follow-up Day 29

On Day 29 (24 hours  $\pm$  1 hour from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment
- AE assessment.

### 8.2.11 Cohort 1: Follow-up Day 30

On Day 30 (48 hours  $\pm$  2 hours from end-of-infusion time on Day 28), the subject will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
- Concomitant medication assessment
- AE assessment

### 8.2.12 Cohort 1: Follow-up Day 33

On Day 33 (120 hours  $\pm$  4 hours from end-of-infusion time on Day 28), subjects will return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PK sample collection (record collection date and time)
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)
- Photography
- Concomitant medication assessment
- AE assessment

### 8.2.13 Cohort 1: Follow-up Day 42

On Day 42 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Exploratory pemphigus immune response biomarkers
- Concomitant medication assessment
- AE assessment

### 8.2.14 Cohort 1: Follow-up Day 56

On Day 56 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position)
- Serum tetanus antibody and VZV antibody
- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Urine IgG
  - Immunophenotyping
  - Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)
- Photography
- Concomitant medication assessment
- AE assessment

### 8.2.15 Cohort 1: Follow-up Day 84

On Day 84 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Serum tetanus antibody and VZV antibody
- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers

- C3
- AECA
- RNAseq
- Urine IgG
- Exploratory pemphigus immune response biomarkers
- Skin biopsy (optional)
- Photography
- Concomitant medication assessment
- AE assessment

Note: Cohort 1 End-of-Study visit is detailed in Section 8.4.

## 8.3 Cohort 2: Subsequent Treatments to Follow-up

### 8.3.1 Cohort 2: Treatment Days 7, 14, 42, 56, 70, and 84

For Cohort 2 Days 7, 14 (all  $\pm$  1 day), 42, 56, 70, and 84 (all  $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- PK sample collection (collected just prior to the start of the study drug infusion) (*Cohort 2, Days 7, 14, and 84 only*)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - $-\Delta FC\Delta$
  - Exploratory pemphigus immune response biomarkers
- Photography

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

# After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest
- 12-lead ECG (to be obtained in triplicate approximately 5 minutes after the completion of study drug infusion (*Cohort 2, Day 14 only*)
- PK sample collection at 5 minutes and 1 and 2 hours after the completion of study drug infusion; record collection date and time for each PK sample (Cohort 2, Days 7, 14, and 84 only)

## Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

## 8.3.2 Cohort 2: Treatment Day 28

For Cohort 2 Day 28 ( $\pm$  3 days), subjects will return to the clinic and the following procedures are to be performed prior to study drug infusion:

- Complete physical exam
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry; to be measured immediately prior to the infusion
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position)
- Serum tetanus antibody and VZV antibody
- PDAI
- PK sample collection (collected just prior to the start of the study drug infusion)
- Immunogenicity sample collection (collected just prior to the start of study drug infusion)
- PD sample collection (collected just prior to the start of the study drug infusion)
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq
  - Immunophenotyping
  - Exploratory pemphigus immune response biomarkers
- Photography
- HR-Qol (ABQoL, Skindex-29)

### After the preceding procedures and assessments are completed:

- Study drug administration (record date and time of dose of study drug)
- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry will be performed at 15, 30, and 45 minutes after the start of the infusion and at completion of the infusion

## After administration of study drug, the following post treatment procedures and assessments will be performed:

- Vital sign measurements (sitting blood pressure, heart rate, respiratory rate, oral temperature) and pulse oximetry: 30 minutes, 1 hour, and 2 hours following completion of the infusion; abnormal results to be repeated after 5 minutes of rest
- PK sample collection at 5 minutes and 1 and 2 hours after the completion of study drug infusion; record collection date and time for each PK sample
- 12-lead ECG (to be obtained in triplicate approximately 5 minutes after the completion of study drug infusion

### Throughout the study visit, the following assessments will be performed:

- Concomitant medication assessment
- AE assessment

### 8.3.3 Cohort 2: Follow-up Day 112

For Cohort 2 Day 112 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - Exploratory pemphigus immune response biomarkers
- Photography
- Concomitant medication assessment
- AE assessment

# 8.4 All Cohorts: End of Study or Early Termination Visit; Cohort 1, Day 112; Cohort 2, Days 91 and 140

For Cohort 1 Day 112 ( $\pm$  5 days) and Cohort 2 Days 91 and 140 ( $\pm$  5 days), subjects are to return to the clinic and the following procedures are to be performed:

- Complete physical exam
- Vital sign measurements (after 5 minutes of rest; sitting blood pressure, heart rate, respiratory rate, oral temperature): abnormal results to be repeated after 5 minutes of rest
- Clinical safety laboratory tests (hematology, serum chemistry panel, urinalysis)
- Pregnancy test
- 12-lead ECG (to be obtained in triplicate after 5 minutes of rest in the supine position) (Cohort 2, Days 91 and 140 only)
- Serum tetanus antibody and VZV antibody
- PDAI
- Immunogenicity sample collection
- PD sample collection
  - IgG, IgG subtypes (IgG1-4), IgA, IgM
  - CIC
  - Anti-Dsg (1 and 3) antibody titers
  - C3
  - AECA
  - RNAseq (Cohort 1 Day 112; Cohort 2, Day 91 only)
  - Urine IgG (Cohort 1 only)
  - Immunophenotyping (Cohort 2, Day 91 only)
  - Exploratory pemphigus immune response biomarkers
- Photography
- HR-Qol (ABQoL, Skindex-29) (Cohort 2 only)
- Concomitant medication assessment
- AE assessment

**Note**: a subject may choose to terminate participation in the study at any time. Under this circumstance, the subject will be encouraged to return as soon as possible for an early termination visit and to receive assessments otherwise scheduled on Day 112 (Cohort 1) or Day 91 (Cohort 2).

## 9. STUDY RULES

## 9.1 Subject Withdrawal

Every reasonable effort will be made to keep the subject in the study; however, if a subject withdraws from the study, the Investigator should complete and report the reasons for withdrawal as thoroughly as possible. The reason(s) for termination must be clearly documented on the appropriate page of the eCRF.

Subjects who have received at least one SYNT001 dose and withdraw or prematurely discontinue study drug should be encouraged to attend, at a minimum, the early termination (ET) visit Day 112 (Cohort 1) or Day 91 (Cohort 2). Subjects in Cohort 2 will also be encouraged to attend the remaining follow up visits on Days 112 and 140.

If the subject fails to return for these assessments for unknown reasons, every effort (eg, telephone, email, and letter) should be made to contact them.

The reason(s) for a subject's participation in the study may be prematurely discontinued will be documented and include:

- 1. The subject wishes to withdraw from the study.
- 2. Request by a regulatory agency or Institutional Review Board).
- 3. The subject experiences a significant or intolerable AE.
- 4. The subject experiences a significant adverse change in vital signs, physical examination findings, or clinical laboratory parameter.
- 5. The subject has a need for a concomitant medication that is not permitted by the study protocol.
- 6. The subject experiences generalized impairment or mental incompetence that would result in the subject being unable to understand his or her participation in the study.
- 7. If, in the Investigator's medical judgment, further participation would be injurious to the health and well-being of the subject, or is not in the best interest of the subject.
- 8. Administrative reasons, such as subject non-compliance or a major protocol violation.

If at the discretion of the Investigator with consultation with the Medical Monitor, a subject requires a significant increase in dose(s) of anti-pemphigus medication(s) for the management of pemphigus, the subject should be encouraged to attend, at a minimum, the ET visit Day 112 (Cohort 1) or Day 91 (Cohort 2). Subjects in Cohort 2 will also be encouraged to attend the remaining follow up visits on Days 112 and 140.

## 9.2 Subject Replacement

Enrolled subjects withdrawn for a reason other than an AE may be replaced.

## 9.3 Study Discontinuation

The Sponsor has the right to terminate or to stop the study at any time. Reasons for study discontinuation may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other related studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Drug supply issues
- Excessive subject self-withdrawal
- Significant protocol violations (eg, violation of eligibility criteria, dosing errors, missing data for study endpoint analysis)

### 9.4 Lost to Follow-up

All reasonable efforts should be made to contact any subject lost to follow-up during the study to complete assessments and retrieve any outstanding data. If the subject is unreachable after three good faith attempts, at a minimum, the Investigator should follow up with a registered letter requesting contact so safety data may be collected, recorded, and reported (if necessary).

### 9.5 Stopping Rules

### 9.5.1 Dose-Escalation Stopping Rule (Cohort 1)

Dose recommendations will be made by a DEC and will be based on safety and PD evaluations including but not limited to, DLTs, AEs, SAEs, and total IgG levels.

Dose-limiting toxicity (DLT) will be defined generally as severe (Grade 3) AEs occurring in ≥2 subjects that are determined to be clinically significant and considered related to study drug.

If 2 or more subjects at any time in any cohort have Grade 3 AEs that are determined to be clinically significant and considered to be related to study drug, dosing will be halted within that cohort and dose-escalation to a higher dose will not occur. Upon review of the available information, the DEC may reduce the dose by at least 50% prior to enrolling additional subjects.

### 9.5.2 Study Stopping Rule

If any subject at any time experiences a life-threatening AE (Grade 4) that is considered to be related to study drug, any further dosing in all enrolled subjects will be suspended until the Sponsor Medical Lead has evaluated the event and determined the next appropriate course of action. At any time during the study, the study may be discontinued if the Sponsor Medical Lead determines that further drug exposure would pose an undue risk to subjects.

### 9.5.3 Individual Stopping Rule

Dosing for any individual subject will be discontinued (ie, no further study drug will be given to that subject) if the subject experiences any study drug-related SAE or any study drug-related

non-serious AE that, in the judgement of the Investigator (following consultation with the Medical Monitor, if desired) or in the judgement of the Sponsor Medical Lead, suggest that it could be unsafe to administer further study drug to that subject.

Subjects who withdraw from this study due to an AE determined to be related to study drug are to be followed until there is:

- Resolution or stabilization of the AE determined to be related
- The subject is lost to follow-up
- The event is otherwise explained

If there is a persistent AE contributing to discontinuation that is determined to be related to SYNT001, subjects must be followed with appropriate medical management until resolution or stabilization. Refer to Section 10 for more information.

Additionally, a subject will be discontinued from further treatment with study drug, at the discretion of the Investigator with consultation with the Medical Monitor, if they require a significant increase in doses of anti-pemphigus medications for the management of pemphigus.

 Syntimmune, Inc.

### 10. EVALUATION OF SAFETY

### **10.1** Safety Parameters

Subjects will be monitored continuously throughout the treatment and follow-up period for AEs (acute, delayed, and/or cumulative), as well as for changes in clinical status. Parameters measure/assess safety include physical examinations, vital sign measurements (including pulse oximetry), clinical (safety) laboratory tests (hematology, serum chemistries, urinalysis), concomitant medication assessments, and ECG. Clinical and laboratory AEs will be graded using the NCI CTCAE; Version 4.03 (see Appendix 1).

### **10.2** Adverse Events

An AE is defined as any untoward medical occurrence in a clinical trial subject associated with the use of a drug, whether considered drug related or not. An AE can be an unfavorable and unintended sign (eg, an abnormal laboratory value finding), a symptom, or a disease temporally associated with the use of a drug, without judgment as to causality. An AE can arise from use of the drug (eg, use in combination with another drug) and from any route of administration, formulation or dose, including an overdose. An AE also includes, but is not limited to, any clinically significant worsening of a pre-existing condition. Examples include:

- Any sign, symptom, physical finding, or laboratory result that has worsened in nature, severity or frequency compared to baseline
- Reactions from an investigational drug, including those occurring because of an overdose, abuse of the study drug, withdrawal phenomena, sensitivity or toxicity
- Concurrent illness that was not present or worsens in nature, severity, or frequency compared to baseline
- Injury or accident
- Exacerbation of a pre-existing condition

Pregnancy is not considered an AE or SAE; however, any pregnancy complication(s) should be recorded as an AE(s) or SAE(s) (if applicable). Elective abortions without complications should not be regarded as AEs, unless they were therapeutic abortions. Hospitalization for normal delivery of a healthy newborn should not be considered an SAE. If a female subject becomes pregnant during the conduct of the study, the Investigator must notify the Sponsor according to the procedures provided in Section 10.5.4.

Planned hospitalization admissions or surgical procedures for a condition known to exist before the subject signed the informed consent are not an AE and should be recorded as medical history. If the planned hospitalization or procedure is executed as planned and without complication, the record in the subject's medical history is considered complete. However, if the event/condition deteriorates in an unexpected manner during the study or following surgery, it must be reported as an AE according to the procedures provided in Section 10.2.1.

### 10.2.1 Recording an Adverse Event

For data collection, all untoward events that occur after informed consent through the last study visit are to be recorded on eCRFs by the investigational site. All AEs are to be accurately recorded on the **Adverse Event** page of the subject's eCRF. The severity of each AE will be graded using the NCI CTCAE, Version 4.03 (see Appendix 1). The date of onset as well as the end date of the event should be recorded or the event should be entered as "ongoing". In addition, the method used to treat the AE and the outcome of the AE will be noted. The Investigator will assess the relationship of the event to study drug.

## **10.2.2** Assessment of Causality

A medically qualified Investigator must assess the relationship of any AE (including SAEs) to the use of the study drug, as related or not related, based on clinical judgment and using all available information. The causal relationship between the study medication and the AE will be assessed using one of the following categories:

Not Related: Factors consistent with an assessment of Not Related include:

- Temporal relationship is lacking (eg, the event did not occur within a reasonable time frame following administration of the study medication); or
- Other causative factors more likely explain the event (eg, a pre-existing condition, other concomitant treatments).

**Related:** Factors consistent with an assessment of Related include:

- There is a positive temporal relationship (eg, the event occurred within a reasonable time frame following administration of study medication); or
- The AE is more likely explained by the investigational product than by another cause (ie, the AE shows a pattern consistent with previous knowledge of the investigational product or the class of the investigational product)

### 10.2.3 Serious Adverse Events

(Notify Medpace Safety within 24 hours; document on eCRF)

The SAE definition and reporting requirements are in accordance with Title 21 Part Code of Federal Regulations (CFR) 312.32 and the Guidance for Industry and Investigators Safety Reporting Requirements for Investigational New Drug (INDs) and Bioavailability /Bioequivalence Studies.

An AE is considered "serious" if, in the view of either the Investigator or sponsor, it results in any of the following outcomes:

• <u>Death:</u> This includes any death that occurs while the subject is "on study" through the last study visit.

 Syntimmune, Inc.

**Note:** Death is an outcome of an AE and not an AE. The event(s) that caused death (eg, illness, accident) is the SAE. Death due to any other cause(s) must also be reported as an outcome of the reportable SAE.

- <u>Life-threatening adverse drug event:</u> An AE or suspected adverse reaction is considered "life threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.
- <u>Inpatient hospitalization or prolongation of existing hospitalization:</u> an AE that requires admission to a hospital for medical and/or surgical intervention.
- In the absence of an AE, the Investigator should <u>not</u> report hospitalization or prolongation of hospitalization as an SAE, as detailed in the following examples:
  - An elective or previously scheduled surgery for a pre-existing condition that has not deteriorated unexpectedly after initiation of treatment (eg, a previously scheduled ventral hernia repair)
  - Hospitalization or prolongation of hospitalization is needed for a procedure required by the protocol
  - Hospitalization or prolongation of hospitalization is part of routine procedure followed by study center
  - o Hospitalization for survey visits, annual physicals, or planned observation
  - Hospitalization for observation with release within 24 hours (eg, an emergency room visit for hematuria that results in a diagnosis of cystitis and discharge to home on oral antibiotics
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Congenital anomaly/birth defect
- <u>Important medical event:</u> An event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

### 10.2.3.1 Recording a Serious Adverse Event

When the diagnosis of an SAE is known or suspected, the Investigator should record the diagnosis or syndrome as the primary SAE term, rather than as signs or symptoms. Signs and symptoms may then be described in the event description. For example, dyspnea should not be used as an SAE term if the diagnosis, which caused the dyspnea, is known to be malignant pleural effusion.

Death should not be recorded as an SAE, but as an outcome of a specific SAE, unless the event preceding the death is unknown. In the exceptional case where the events leading to death are unknown, then death may be used as an event term. If an autopsy was performed, the autopsy the autopsy report should be provided.

### 10.2.3.2 Reporting a Serious Adverse Event

#### RESPONSIBILITIES OF THE INVESTIGATOR

Any death, SAE, or pregnancy, experienced by the subject after informed consent through the last study visit, regardless of relationship to study drug, must be promptly reported (within 24 hours of the Investigator becoming aware of the event) by telephone or electronic transmission to the Sponsor (or designee).

Contact information for SAE reporting:



Additionally, the Investigator will be able to contact the **Medical Monitor**:

## **Medical Safety Contact**



The Investigator will report the SAE to his or her IRB in accordance with IRB's standard operating procedures and policies. Adequate documentation must be maintained showing that the IRB was properly notified.

SAEs must be recorded on the SAE form in the electronic data capture (EDC) system. This requirement includes all SAEs that occur after informed consent through the last study visit. The minimum information required for SAE reporting includes identity of investigator, site number, subject number, an event description, SAE term(s), onset date, the reason why the event is serious (ie, the seriousness criteria), and the Investigator's assessment of the relationship of the event to study treatment. Additional SAE information including medications or other therapeutic measures used to treat the event, action taken with the study treatment due to the event, and the outcome/resolution of the event will be recorded. Paper forms for reporting SAEs will be provided to the study sites as back-up in case the EDC system is not accessible.

In all cases, the Investigator should continue to monitor the clinical situation and report all material facts relating to the progression or outcome of the SAE. Furthermore, the Investigator may be required to provide supplementary information as requested by the Sponsor (or designee).

### RESPONSIBILITIES OF THE SPONSOR (OR DESIGNEE)

The Sponsor (or designee) will process and evaluate all SAE as soon as the reports are received. For each SAE received, the Sponsor will decide as to whether the criteria for expedited reporting have been met.

The Sponsor (or designee) is responsible for promptly informing the FDA and other regulatory authorities as well as other participating Investigators of the event. Written submission must be made by the Sponsor to the FDA as soon as possible and in no event later than 15 calendar days after the Sponsor's initial notification of the event, or for an event that is fatal or life-threatening no later than 7 calendar days after the Sponsor's initial notification.

### EXPEDITED REPORTING

Under FDA ruling (US Code of Federal Regulations, Title 21 CFR Part 312.32) and the ICH Guideline "Clinical Safety Data Management: Definitions and Standards for Expedited Reporting E2A," the Sponsor is required to submit written documentation, in the form of a safety report, detailing:

- Any event associated with the use of the drug, that is both serious and unexpected, or
- Any finding from tests in laboratory animals that suggests a significant risk for human subjects, including reports of mutagenicity, teratogenicity, or carcinogenicity.

The Sponsor will submit SAEs that meet the criteria for expedited reporting to the regulatory authorities in accordance with local regulations governing safety reporting.

### 10.2.4 Follow-Up of Adverse Events and Serious Adverse Events

Any SAE or AE must be followed until either resolution of the event or determination by the Investigator that the event has become stable or irreversible. Appropriate diagnostic tests should be performed and therapeutic measures, if indicated, should be instituted until the event has returned to baseline or until a clinically satisfactory resolution has been achieved. The appropriate follow-up visits must be scheduled and the specific tests repeated or performed as necessary. The status of all AEs will be documented as of the last study visit. If all required information is not available at the time of the initial report, follow-up information will be completed in the EDC system.

### **10.3** Warnings and Precautions

#### 10.3.1 Vaccinations

Subjects must not receive any vaccinations from within 2 weeks of screening until 28 days following final dose of study drug.

## 10.3.2 Management of Allergic or Infusion-Related Reactions

As observed with all mAbs administered by IV infusion, infusion-related reactions to SYNT001 are possible. In general, infusion reactions to mAbs observed in human studies typically develop

 Syntimmune, Inc.

within 30 minutes to 2 hours after the initiation of drug infusion, although symptoms may be delayed for up to 24 hours. These infusion reactions can occur with the first dose of a mAb and are generally mild in severity, although severe and even fatal reactions can occur.

Allergic and/or infusion-related reactions include hypersensitivity reactions and cytokine release syndromes. These reactions are experienced by subjects during or within hours of the infusion of mAb therapy. Symptoms can include flushing, alterations in heart rate and blood pressure, dyspnea, bronchospasm, back pain, fever, urticaria, edema, nausea, and all types of rashes. Anaphylaxis is recognized as a severe, life-threatening, generalized, or systemic reaction. This is a medical emergency characterized by rapidly developing life-threatening airway and/or breathing and/or circulation problems usually associated with skin or mucosal changes.

Management of Grade 1 infusion reactions include interrupting the infusion or decreasing the rate of infusion by 50% and observing. Symptoms may also be treated as needed with medications such as diphenhydramine, hydrocortisone, or acetaminophen, either alone or in combination, depending on the subject's signs and symptoms. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 preparation.

Management of Grade 2 and higher infusion reactions should include stopping the infusion of study drug. Continued treatment with SYNT001 is prohibited following Grade 2 or higher infusion reactions. See Figure 2 and Figure 3 for details on the management of Grade 2 and Grade 3 infusion reactions. Allergic or IRRs will be graded in severity and managed based on NCI CTCAE Version 4.03 (see Table 8).

Figure 2. Management of Moderate (Grade 2) Infusion Reactions



If symptoms and signs resolve completely either spontaneously or after administration of diphenhydramine with or without hydrocortisone, consider rechallenge:

Wait at least 20 minutes following medication administration before commencing rechallenge at an infusion rate of 50% or less of the initial infusion rate or

Consider pre-medicating the subject with the same medication(s) 20-30 minutes in advance of subsequent administrations of SYNT001 and starting infusion at 50% of the planned infusion rate for the first 30 minutes, then returning to the intended infusion rate in the absence of any infusion reaction. If the infusion is interrupted or the infusion rate is decreased, it is important to note that all study drug infusions must be completed within 4 hours of SYNT001 administration.
Figure 3. Management of Severe (Grade 3 or Higher) Infusion Reactions

Subject presents with any of the below:

- Urticaria
- Airway threatened by angioedema
- Angioedema: Lip, mouth, facial swelling
- Respiratory compromise wheezing, dyspnea, stridor or hypoxia (O<sub>2</sub> saturation <90%)</li>
- BP <90 mmHg SBP or >30% decrease from patient baseline



### Start basic life support:

- High oxygen flow
- On bed, head down, legs up
- Large bore IV cannula, 1 L normal saline STAT
- Initiate vital signs at least every 15 minutes



Consider (under medial direction):

Epinephrine 1:1000

• 0.3 mg (0.3 mL) IM into lateral thigh



Airway Threatened: Nebulized epinephrine 1:1000, 3–5 mL (3–5 mg)

**Bronchospasm:** Nebulized salbutamol 5 mg

(Wheeze or Hypoxia) Consider: Intubation / nebulized epinephrine

**Hypotension:** Place on cardiac monitor

(Systolic BP <100 mmHg) Further epinephrine 1:1000, 0.3 mg IM and

IV normal saline bolus 20 mL/kg STAT as needed

Have vasopressin on hand



Transfer to Emergency Room/ICU Observe until all symptoms resolved.

 Table 8.
 Grading and Management of Allergic or Infusion-Related Reactions

| Adverse | | | Grade | | |
|---|---|---|---|---|---|
| Event | 1 | 2 | 3 | 4 | 5 |
| Infusion-<br>related<br>reaction | Mild transient<br>reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, nonsteroidal antiinflammatory drugs [NSAIDS], narcotics, IV fluids): prophylactic medications indicated for ≤24 hours | Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Allergic<br>reaction | Transient<br>flushing or<br>rash, drug<br>fever<br><38.0°C.<br>Intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤24 hours | Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (eg, renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Anaphylaxis | _ | _ | Symptomatic<br>bronchospasm, with or<br>without urticarial;<br>parenteral intervention<br>indicated; allergy-related<br>edema/angioedema;<br>hypotension | Life-<br>threatening<br>consequences;<br>urgent<br>intervention<br>required | Death |
| Cytokine<br>release<br>syndrome | Mild reaction;<br>infusion<br>interruption<br>not indicated;<br>intervention<br>not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (eg, antihistamines, NSAIDS, narcotics, IV fluids): prophylactic medications indicated for ≤24 hours | Prolonged (eg, not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement, hospitalization indicated for clinical sequelae (eg, renal impairment, pulmonary infiltrates) | Life-<br>threatening<br>consequences;<br>pressor or<br>ventilator<br>support<br>indicated | Death |

Abstracted from NCI CTCAE Version 4.03.

### **10.3.3** Potential Immune Effects

An antibody blocking FcRn is anticipated to have several effects. These include acceleration of catabolism of IgG, but not other immunoglobulin isotypes such as IgA and IgM, leading to dose-dependent decreases in circulating IgG levels by up to an estimated 50% from the baseline levels

after a single dose and further decreases after multiple doses up to a 70% to 80% reduction. Based on studies in humans, it is expected that with a single dose, the nadir of this effect will occur approximately 5 days after dosing. The time course of recovery of IgG following dosing in the Phase 1a study suggests that a return to within 30% of baseline levels observed at pretreatment occurs within 4 weeks after a single dose and within 4 weeks after multiple doses as shown in NHPs.

Given the normal adult range of total IgG of 500 to 1600 mg/dL (Agarwal and Cunningham-Rundles, 2007; Furst, 2009; Gonzalez-Quintela et al., 2008; Jolliff et al., 1982; Keystone et al., 2007; McMillan et al., 1997; van Vollenhoven et al., 2013), with a mean of 1150 mg/dL, a 50% decrease in mean total IgG would translate to 575 mg/dL and a 50% decrease from the low end of the normal range used for the inclusion criteria of 600 mg/dL in this study would be to 300 mg/dL. An 80% decrease from baseline after multiple doses would result in IgG levels of 230 mg/dL and 120 mg/dL, respectively. While these levels are in the range found in patients with primary humoral immunodeficiency (Ameratunga et al., 2013), the levels will be transient. Further, as reported for other therapies used for pemphigus, the temporary (ie, less than 4 months) depletion of IgG (up to 95% reduction of total IgG as seen with immunoadsorption) does not appear to impart an increased risk of infection (Eming and Hertl, 2006; Furst, 2009; Keystone et al., 2007; Schmaldienst et al., 2001; van Vollenhoven et al., 2013). Study subjects will be monitored clinically for any infection. Further, commercial IVIG can be given to immediately restore IgG levels in case of a bacterial infection occurring while their IgG levels are decreased.

An antibody that blocks FcRn is expected to also down-modulate innate and adaptive immunity and the catabolism of IgG-containing ICs. Specifically, it is expected that anti-FcRn will promote the clearance of IgG-containing ICs and the effects of these ICs on stimulating innate immune cell production of inflammatory cytokines (eg, interleukin 12 [IL-12], interferon-γ, and tumor necrosis factor) and inhibit the processing and presentation of antigens contained within ICs and thus the antigen-specific activation of CD4<sup>+</sup> and CD8<sup>+</sup> T-cells. Therefore, subjects with pre-existing conditions that are dependent upon IgG antibodies, such as chronic infections (eg, HIV, hepatitis B virus [HBV] or hepatitis C virus [HCV]), will be excluded from this study, as will subjects with active infection, in general.

### **10.4** Events of Special Interest

Not applicable.

### 10.5 Other Safety Considerations

### 10.5.1 Laboratory Data

All laboratory data obtained during the study should be reviewed. Any abnormal value that leads to a change in subject management (eg, requirement for additional medication or monitoring) or is determined to be of clinical significance by the Investigator should be reported as an AE and/or SAE as appropriate, unless this value is consistent with values obtained before entry into the study.

 Syntimmune, Inc.

### **10.5.2 Medication Errors**

Any medication error that results in an AE, even if it does not meet the definition of serious, requires reporting within 24 hours to the safety Medical Monitor. Refer to Section 10.2.3.2 for more information.

### **10.5.3 Overdose**

For the purposes of this study, an overdose of SYNT001 is defined as a dose that is two-fold higher than the intended dose for the subject. As all dosing for this study will be conducted in a controlled clinical setting, an overdose is not anticipated. In the unlikely event an overdose should occur, it should be reported as an AE.

### 10.5.4 Pregnancy

If a female subject or the female partner of a male subject becomes pregnant during the course of the study, the Investigator must report the pregnancy to Medpace Safety using the **Pregnancy Reporting Form** within **24 hours** of becoming aware of the event. The Investigator must obtain consent to collect pregnancy information (including the status of the newborn, if applicable).

If some of the information required for completion of the Pregnancy Reporting Form is unavailable at the time of the initial report, follow-up reports will be completed and submitted within 24 hours of becoming aware of the new information. Any pregnancy will be followed through delivery for the observation of any SAEs. Any SAE that occurs during pregnancy must be recorded on the SAE report form in the EDC system (eg, maternal serious complications, therapeutic or spontaneous abortion, ectopic pregnancy, stillbirth, neonatal death, congenital abnormality, birth defect) and reported within 24 hours in accordance with the procedure for reporting SAEs (see Section 10.2.3.2).

### 11. STATISTICAL CONSIDERATIONS

### 11.1 General Design

This study is being conducted to evaluate the safety, tolerability, PK, PD, activity, and immunogenicity of SYNT001 in pemphigus patients.

### 11.2 Study Populations

Three populations will be employed in the analysis of study data:

- The Safety population will consist of all subjects who have received at least one dose of study drug.
- The **PD** population will consist of all subjects who receive at least one dose of study drug and have post-dose PD data available.
- The **PK** population will consist of all subjects who receive at least one dose of study drug and have post-dose PK data available.

Primary safety analyses will be performed on the Safety population. Demographics, subject disposition, screening, and baseline characteristics will be summarized for the Safety, PK, and PD populations, where appropriate.

### 11.3 Sample Size Justification

Formal sample size calculations were not performed. The number of subjects was chosen based on feasibility and was considered sufficient to meet the study objectives.

### 11.4 Statistical Analysis

### 11.4.1 Statistical Analysis Plan

Detailed methodology for summary and statistical analyses of the data collected in this study will be documented in a statistical analysis plan (SAP). The SAP may modify the plans outlined in the protocol; however, any deviations from the previously approved statistical plan will be described and justified in a SAP amendment. Additional statistical analyses other than those described in this section may be performed if deemed appropriate and will be described in the SAP. The SAP will be finalized prior to database lock.

Statistical analyses will be performed using Statistical Analysis System (SAS) software version 9.4 or later (Cary, NC). All clinical data captured will be provided in data listings.

Methods of handling of missing data for different endpoints will be further specified in the SAP. In general, where individual data points are missing because of insufficient samples, dropouts, or other reasons, the data will be analyzed based on reduced denominators unless specified otherwise in the SAP.

# 11.4.2 Statistical Methodology

All clinical data captured will be provided in data listings. Subject disposition, demographic information, and baseline characteristics will be presented. Baseline will be defined at the last value obtained prior to the first dose of study drug. Results will be summarized by dose level and cohort. Any discrepancy between treatment to be given and treatment received will be accounted for in these displays.

Continuous data will be summarized using descriptive statistics: number of subjects (N), number of observations (n), mean, median, standard deviation (SD), minimum, and maximum.

Categorical data will be summarized using frequencies and percentages. When categorical data will be presented, the percent will be suppressed when the count is zero to draw attention to the non-zero counts. The denominator for all percentages, unless otherwise specified, will be the number of subjects in the specified analysis population.

### 11.4.3 Analysis of Primary Endpoints

### 11.4.3.1 Safety Analysis

All statistical analysis of safety outcomes will be descriptive. The evaluation of SYNT001 based on vital signs, physical examination, ECGs, clinical safety laboratory tests, the incidence of AEs, TEAEs, and SAEs will be summarized by dose and dose regimen, severity, and relationship to study drug.

TEAEs will be summarized using the Medical Dictionary for Regulatory Activities (MedDRA®; Version 19 or higher) System Organ Class (SOC) and preferred term, classified from verbatim terms. The incidence and percentage of subjects with at least one occurrence of a preferred term will be included, using the most severe grade. The number of events per preferred term will also be summarized. Causality (relationship to study drug [related/not related]) will be summarized separately.

TEAEs, SAEs, and AEs leading to withdrawal, dose modification, or treatment discontinuation will be listed by subject per SOC and preferred terms. Duration of AEs will be determined and included in listings, along with action taken and outcome.

Laboratory results will be summarized by visit, time point, dose, and dose regimen. The incidence of laboratory abnormalities will be summarized. The worst on-study grade after the first dose of study drug will be summarized. Results for variables that are not coded will be presented in the listings as below, within, and above the normal limits of the central laboratory.

Vital sign measurements and change from baseline will be summarized at each scheduled time point by cohort using descriptive statistics.

Arithmetic mean of parameters from triplicate ECG will be calculated first for each subject at each planned time point. Then summary statistics of ECG test parameters (mean of triplicate) and change from baseline to each post-dose time point will be calculated. Shift tables for ECG test result category change (normal, abnormal, clinically abnormal) from pre-dose to each post-

 Syntimmune, Inc.

dose time point showing number and percentage of subjects with movement between categories will be presented by treatment group. Frequency and percentage of subjects experiencing potential QTc prolongation (QTcF > 450) will be summarized at each time point by cohort.

Concomitant medications will be coded using WHO Drug Dictionary (WHO-DD March 2013, Type B2 or later) and the data will be summarized and presented in tables and listings.

### 11.4.3.2 Dose Selection Data

The evaluation of SYNT001 based on total IgG levels and responses on the PDAI total activity score from baseline will be summarized using descriptive statistics. Descriptive statistics will include mean, SD, coefficient of variation (CV), median, minimum, and maximum. The determination of dose and dosing duration of SYNT001 that achieves (i) total IgG level nadir decrease by  $\geq$ 60% and  $\leq$ 90% from baseline and (ii) a PDAI total activity score of  $\geq$ 50% reduction from baseline to allow further clinical development in subject with pemphigus (vulgaris or foliaceus).

### 11.4.4 Analysis of Secondary Endpoints

### 11.4.4.1 Pharmacokinetic Analysis

PK results for SYNT001 will be summarized by dose and dose regimen, visit and time point.

Descriptive statistics will be provided for the PK parameters including mean, SD, CV, median, minimum, and maximum.

For calculation of mean concentrations and generation of mean concentration-time profiles, all below the limit of quantification (BLQ) values will be set to zero except when an individual BLQ falls between 2 quantifiable values, in which case it will be omitted.

If there are values above the BLQ, but too sparse to allow full analysis, descriptive statistics will be performed on available values.

### 11.4.4.2 Pharmacodynamic Analysis

Disease activity marker results will be summarized by dose, dose regimen and visit. Descriptive statistics of PD will include mean, SD, median, minimum, and maximum.

### 11.4.4.3 Immunogenicity Analysis

Immunogenicity results will be summarized by cohort, visit and time point. Descriptive statistics will include mean, SD, CV, median, minimum, and maximum.

### 11.4.4.4 PDAI Data

PDAI results will be summarized by score (total activity score, total damage score), cohort, and visit. Descriptive statistics will include absolute change from baseline, and percent change from

 Syntimmune, Inc.

baseline. PDAI will also be summarized by disease severity category, mild (0 to 8), moderate (9 to 24), and severe ( $\geq$ 25).

### 11.4.5 Analysis of Exploratory Endpoints

### 11.4.5.1 Corticosteroid Use

The evaluation of corticosteroid use during the study will be summarized by dose, dose regimen and visit.

# 11.4.5.2 Health-Related Quality of Life Data

HR-QoL results from the ABQoL and Skindex-29 assessments will be summarized by dose, dose regimen, and visit.

# 11.4.5.3 Photography

The qualitative assessment of changes in appearance of skin and mucosal lesions as determined by photography presented by dose, dose regimen, and visit.

# 11.5 Interim Analysis

No interim analysis is planned.

### 12. STUDY MANAGEMENT

### 12.1 Regulatory and Ethical Considerations

### 12.1.1 Ethical Conduct

The study must fully adhere to the principles outlined in "Guideline for Good Clinical Practice" ICH E6 Tripartite Guideline (January 1997), and in general, be conducted in a manner consistent with the principles described in the Declaration of Helsinki. The Investigator will ensure that the conduct of the study complies with the basic principles of GCP as outlined in the current version of 21 CFR, subpart D, Part 312, "Responsibilities of Sponsors and Investigators", Part 50, "Protection of Human Subjects", and Part 56, "Institutional Review Boards".

### 12.1.2 Informed Consent

A signed informed consent form (ICF) in compliance with 21 CFR, Part 50.25(a) and Part 50.25(b) and the ICH guidelines, will be obtained from each subject before the subject is entered into the study and before any study screening procedure is performed that involves risk. The method of obtaining and documenting the informed consent will comply with ICH GCP and all applicable laws and regulations and will be subject to approval by the Sponsor.

The Investigator, or designee, is responsible for obtaining written informed consent from each subject (or the subject's legally authorized representative) participating in this study after a thorough and clear explanation of the objectives, procedures, anticipated benefits, and potential hazards of the study. In the case where the subject is unable to read, an impartial witness should be present during the entire informed consent discussion. After the subject has orally consented to participation in the trial, the witness' signature on the form will attest that the information in the consent form was accurately explained and understood. The study site must retain the original ICF and a copy must be provided to the subject or to the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

The Sponsor, or designee, must review the signed ICF against any proposed deviations from a sample ICF the Sponsor has supplied to each site. The final IRB-approved document must be provided to the Sponsor for regulatory purposes.

The eCRF for this study contains a section for documenting informed subject consent, and this must be completed appropriately. Signed ICFs must remain in each subject's study file and must be available for verification by site monitors at any time. If new safety information results in significant changes in the risk/benefit assessment, the consent form should be reviewed and updated as necessary. All subjects (including those already being treated) should be informed of the new information, should be given a copy of the revised form, and should give their consent to continue in the study.

### 12.1.3 Subject Confidentiality and Privacy

As applicable, in accordance with the Health Insurance Portability and Accountability Act (HIPAA), and associated privacy regulations, a patient authorization to use personally

 Syntimmune, Inc.

identifiable health information may be required from each patient before research activities begin.

The Investigator must ensure that subjects' anonymity will be maintained and that their identities are protected from unauthorized parties. On eCRFs or other documents submitted to the Sponsor, subjects should be identified by an identification code and not by their names. The Investigator should keep a subject enrollment log showing codes, names, and addresses. The Investigator should maintain documents intended for storing onsite (eg, subjects' written consent forms) in strict confidence.

All study drugs, subject bodily fluids and tissue, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by the Sponsor.

### 12.1.4 Future Use of Stored Specimens

Not all the tissue and blood components obtained during this study may be required for the tests that are part of the clinical trial. Available samples may be used for additional analyses and research. This research will help to understand disease subtypes, drug response, and AEs, and possibly identify new drug targets or biomarkers that predict subject response to treatment. The use of the samples for internal research will adhere to the guidelines defined by the FDA in "Guidance on Informed Consent for In Vitro Diagnostic Device Studies Using Leftover Human Specimens that are Not Individual Identifiable" (issued 25 April 2006) and the European Medicines Agency "Reflection Paper on Pharmacogenetic Samples, Testing and Data Handling" (Doc. Ref. EMEA/CHMP/PGxWP/201914/2006; 15 November 2007). If a subject requests destruction of their tissue and blood samples and the samples have not yet been de-identified, the Sponsor will destroy the samples as described in the FDA guidance. The Sponsor will notify the Investigator in writing that the samples have been destroyed.

### 12.2 Study Administration

The study administration structure is provided in Table 9.





# 12.2.1 Institutional Review Board Approval

This study is being conducted under US IND 132727. This protocol (and any modifications) and appropriate consent procedures must be reviewed and approved by the site-specific IRB before the study is initiated. The IRB must operate in accordance with the current federal or local regulations. The Investigator will send a letter or certificate of IRB approval to the Sponsor (or designee) before subject enrollment and whenever subsequent modifications to the protocol are made.

### 12.2.2 Data Handling and Record Keeping

All data will be entered in a validated electronic data capture system using single data entry. Standard procedures (including following data review guidelines, manual clinical review based on subject profiles, computerized validation to produce queries, and maintenance of an audit file, which includes all database modifications) will be followed to ensure accurate data. Clinical personnel will review all data listings for outliers, data inconsistencies, and spelling errors.

### 12.2.3 Data Protection

The Investigator agrees that all information received from the Sponsor, including but not limited to the IB, this protocol, eCRFs, the INDs, and any other study information remain the sole and exclusive property of the Sponsor during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) or otherwise into the public domain without prior written consent from the Sponsor.

### 12.2.4 Study Site Regulatory Documentation

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should

be classified into 2 separate categories as follows: (1) Investigator's study file and (2) subject clinical source documents (see Section 12.2.5).

The Investigator's study file will contain the protocol and protocol amendments, eCRFs, query forms, IRB and governmental approval with correspondence, sample informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

Subject clinical source documents (usually predefined by the project to record key efficacy and safety parameters independent of the eCRFs) may include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, electroencephalogram, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject screening and enrollment logs. The Investigator must keep these two categories of documents on file for at least 2 years following the marketing application approval date for the study treatment and for the indication being investigated or for 2 years after the development program is discontinued and the FDA notified. After that period, the documents may be destroyed subject to local regulations with prior written permission from the Sponsor. If the Investigator wants to assign the study records to another party or move them to another location, the Sponsor must be notified in advance.

If the Investigator cannot guarantee the archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and the Sponsor to store these in a sealed container outside of the study site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storing outside of the study site.

### 12.2.5 Subject Clinical Source Documents and Background Data

Investigators must maintain adequate and accurate source documents on which the eCRFs for each subject are based. They are separate and distinct from the eCRFs.

These records include detailed notes on the following:

- Medical history
- Informed consent
- HIPAA authorization, if applicable (either contained in the ICF or presented to the subject candidate as a standalone document)
- Description of the complete consenting process
- The basic identifying information that linked the subject's medical record with the eCRFs
- The results of all diagnostic tests performed, diagnoses made, therapy provided, and any other data on the condition of the subject
- The medical condition of the subject during their involvement in the study
- All AEs
- The subject's exposure to the study medication
- The subject's exposure to any concomitant therapy
- All relevant observations and data on the condition of the subject throughout the trial
- Justification for all entries in the subject's eCRF

A subject log of all potentially eligible subjects considered, but not consented, for obvious deviations from the entry criteria, will be kept at each site. The log will contain subjects' initials, diagnosis, eligibility, or, if not eligible, reason for not consenting. All consented subjects will be logged, regardless of whether they ultimately enroll.

Upon request, the Investigator will supply the Sponsor with any required background data from the study documentation or clinic records. This is particularly important when eCRFs are illegible or when errors in data transcription are suspected. In case of special problems or governmental queries or requests for audit inspections, it is also necessary to have access to the complete study records, provided that subject confidentiality is protected.

### 12.2.6 Electronic Case Report Forms

Clinical trial data for this study will be captured on eCRF designed for computer processing and analysis. This computerized system will be validated and compliant with 21 CFR Part 11, as described in the FDA guidance "Use of Electronic Records and Electronic Signatures in Clinical Investigations Under 21 CFR Part 11 – Questions and Answers." If corrections are made after review and sign-off by the Investigator, he/she must be aware of the changes and provide written acknowledgement. There will also be an electronic audit trail. Corrections on paper CRFs must be initialed and dated by the person making the change. The Investigator agrees to provide all information requested on the eCRF in an accurate manner using instructions provided. The Investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported to the Sponsor in the eCRF and in all required reports.

An eCRF is required to be submitted for every subject who receives any amount of study drug. This includes submission of retrievable data on subjects who withdraw before completion of the study. Prior to submission, eCRFs must be reviewed for completeness and accuracy, and signed and dated where indicated, by the Investigator or designee. If a subject stops treatment or terminates from the study, the dates and reasons must be noted on the eCRF.

# 12.3 Clinical Monitoring, Audits, and Inspections

The Investigator and study staff are responsible for maintaining a comprehensive and accurate filing system of all study-related documentation that will be suitable for inspection for routine monitoring, audit, or inspection at any time by the Sponsor (or designee) and/or a regulatory authority.

### 12.3.1 Clinical Monitoring

During the clinical study, it is understood that the responsible Sponsor site monitor or designee (eg, contract research organization [CRO]) will contact and visit the study site at regular intervals for routine monitoring of various records. Routine monitoring activities will be conducted to verify adherence to the protocol, completeness, consistency and accuracy of the data, and to review study source documents and drug accountability records. Regular review of the eCRFs for completeness, clarity, and to cross-check against source documents is required to

 Syntimmune, Inc.

monitor the progress of the study. Data will be reviewed and verified against the source documents (eg, original medical records and laboratory results) to ensure validity.

The Investigator will provide the Sponsor or designee with full access to all source data (including laboratory tests) and provide administrative support if requested. The Investigator (or designee) must agree to cooperate with the site monitor to ensure that any problems detected during these monitoring visits are resolved.

Site-specific study procedures, such data-recording and handling of the data, may be assessed during the study by a Clinical Quality Assurance representative(s) authorized by the Sponsor. Further, this designee, as well as the site monitor, will be permitted to inspect the study documents (study protocol, eCRFs, study drug accountability, original study-relevant medical records) to ensure that the study is conducted in compliance with the protocol.

During these visits, all representatives of the Sponsor will be responsible for ensuring data integrity and subject confidentiality is protected.

### 12.3.2 Audits and Inspections

Clinical site and study audits will be conducted as necessary to assure the validity of the study data. The Sponsor (or designee) may perform a quality assurance audit to ensure compliance with GCP, this protocol, and all applicable regulatory requirements. The Investigator should ensure that study documents (protocol, eCRFs, study drug record-keeping, original study-relevant medical records) are made available to the Sponsor (or designee) for examination. All subject data will be treated as confidential.

A regulatory authority, after appropriate notification, may also wish to conduct an inspection during the study or even after its completion. If a regulatory authority requests an inspection, the Investigator must immediately inform the Sponsor.

### 12.4 Changes to the Protocol

Protocol modifications to ongoing studies must be made only after consultation between a Sponsor representative and the Investigator. Protocol modifications will be prepared, reviewed, and approved by Sponsor representatives.

All protocol modifications must be submitted to the IRB for information and approval in accordance with local requirements, and to regulatory agencies, if required. Approval must be obtained before any changes can be implemented, except for changes necessary to eliminate an immediate hazard to study subjects, or when the change involves only logistical or administrative aspects of the trial (eg, change in site monitor, change of telephone number).

### 12.5 Study Discontinuation and Closure

The Sponsor has the right to terminate the study at any time. In terminating the study, the Sponsor and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests.

 Syntimmune, Inc.

### 13. PUBLICATION AND DATA SHARING POLICY

The results of this study may be published or presented at scientific meetings. The Investigator agrees that any manuscript or abstract they author may be published only after receiving written permission from the Sponsor.

If the Sponsor coordinates a publication or presentation of study results from all study sites, the participation of Investigator or other representatives of study site as a named author shall be determined in accordance with the Sponsor's policy and generally accepted standards for authorship as developed by the International Committee of Medical Journal Editors (ICMJE) and in accordance with Good Publication Practices.

### 14. REFERENCES

Agarwal S, Cunningham-Rundles C. Assessment and clinical interpretation of reduced IgG values. Ann Allergy Asthma Immunol. 2007;99(3):281-3.

Ameratunga R, Woon ST, Gillis D, Koopmans W, Steele R. New diagnostic criteria for common variable immune deficiency (CVID), which may assist with decisions to treat with intravenous or subcutaneous immunoglobulin. Clin Exp Immunol. 2013;174(2):203-11.

Blaha M, Pitha J, Blaha V, Lanska M, Maly J, Filip S, et al. Experience with extracorporeal elimination therapy in myasthenia gravis. Transfus Apher Sci. 2011;45(3):251-6.

Chren MM, Lasek RJ, Quinn LM, Mostow EN, Zyzanski SJ. Skindex, a quality-of-life measure for patients with skin disease: reliability, validity, and responsiveness. J Invest Dermatol. 1996;107(5):707-13.

Eming R, Hertl M. Immunoadsorption in pemphigus. Autoimmunity. 2006;39(7):609-16.

Furst DE. Serum immunoglobulins and risk of infection: how low can you go? Semin Arthritis Rheum. 2009;39(1):18-29.

Gonzalez-Quintela A, Alende R, Gude F, Campos J, Rey J, Meijide LM, et al. Serum levels of immunoglobulins (IgG, IgA, IgM) in a general adult population and their relationship with alcohol consumption, smoking and common metabolic abnormalities. Clin Exp Immunol. 2008;151(1):42-50.

Hsu DY, Brieva J, Sinha AA, Langan SM, Silverberg JI. Comorbidities and inpatient mortality for pemphigus in the U.S.A. Br J Dermatol. 2016;174(6):1290-8.

Jolliff CR, Cost KM, Stivrins PC, Grossman PP, Nolte CR, Franco SM, et al. Reference intervals for serum IgG, IgA, IgM, C3, and C4 as determined by rate nephelometry. Clin Chem. 1982;28(1):126-8.

Kasperkiewicz M, Ellebrecht CT, Takahashi H, Yamagami J, Zillikens D, Payne AS, et al. Pemphigus. Nat Rev Dis Primers. 2017;3:17026.

Keystone E, Fleischmann R, Emery P, Furst DE, van Vollenhoven R, Bathon J, et al. Safety and efficacy of additional courses of rituximab in patients with active rheumatoid arthritis: an open-label extension analysis. Arthritis Rheum. 2007;56(12):3896-908.

Kohler W, Bucka C, Klingel R. A randomized and controlled study comparing immunoadsorption and plasma exchange in myasthenic crisis. J Clin Apher. 2011;26(6):347-55.

Langan SM, Smeeth L, Hubbard R, Fleming KM, Smith CJ, West J. Bullous pemphigoid and pemphigus vulgaris--incidence and mortality in the UK: population based cohort study. BMJ. 2008;337:a180.

McMillan SA, Douglas JP, Archbold GP, McCrum EE, Evans AE. Effect of low to moderate levels of smoking and alcohol consumption on serum immunoglobulin concentrations. J Clin Pathol. 1997;50(10):819-22.

Nixon AE, Chen J, Sexton DJ, Muruganandam A, Bitonti AJ, Dumont J, et al. Fully human monoclonal antibody inhibitors of the neonatal fc receptor reduce circulating IgG in non-human primates. Front Immunol. 2015;6:176.

Roopenian DC, Christianson GJ, Sproule TJ, Brown AC, Akilesh S, Jung N, et al. The MHC class I-like IgG receptor controls perinatal IgG transport, IgG homeostasis, and fate of IgG-Fc-coupled drugs. J Immunol. 2003;170(7):3528-33.

Rosenbach M, Murrell DF, Bystryn JC, Dulay S, Dick S, Fakharzadeh S, et al. Reliability and convergent validity of two outcome instruments for pemphigus. J Invest Dermatol. 2009;129(10):2404-10.

Schmaldienst S, Mullner M, Goldammer A, Spitzauer S, Banyai S, Horl WH, et al. Intravenous immunoglobulin application following immunoadsorption: benefit or risk in patients with autoimmune diseases? Rheumatology. 2001;40(5):513-21.

Sebaratnam DF, Hanna AM, Chee SN, Frew JW, Venugopal SS, Daniel BS, et al. Development of a quality-of-life instrument for autoimmune bullous disease: the Autoimmune Bullous Disease Quality of Life questionnaire. JAMA Dermatol. 2013;149(10):1186-91.

Sebaratnam DF, Okawa J, Payne A, Murrell DF, Werth VP. Reliability of the autoimmune bullous disease quality of life (ABQOL) questionnaire in the USA. Qual Life Res. 2015;24(9):2257-60.

Shimizu T, Takebayashi T, Sato Y, Niizeki H, Aoyama Y, Kitajima Y, et al. Grading criteria for disease severity by pemphigus disease area index. J Dermatol. 2014;41(11):969-73.

van Vollenhoven RF, Emery P, Bingham CO, 3rd, Keystone EC, Fleischmann RM, Furst DE, et al. Long-term safety of rituximab in rheumatoid arthritis: 9.5-year follow-up of the global clinical trial programme with a focus on adverse events of interest in RA patients. Ann Rheum Dis. 2013;72(9):1496-502.

# APPENDIX 1. NCI CTCAE, VERSION 4.03

 Syntimmune, Inc.

# Common Terminology Criteria for Adverse Events (CTCAE)

# Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

### Common Terminology Criteria for Adverse Events v4.0 (CTCAE) Publish Date: May 28, 2009

### Quick Reference

The NCI Common Terminology Criteria Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

### **Components and Organization**

### SOC

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e. SOC Investigations for laboratory test results). CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

### **CTCAE Terms**

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disea temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analysis Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

# Definitions

A brief definition is provided to clarify the meaning of each AE term.

### Grades

displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic telephone, managing money, etc. observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated; medications, and not bedridden. limiting age-appropriate instrumental ADL\*.

Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL\*\*.

Grade 4 Life-threatening consequences; urgent intervention indicated.

Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than e options for Grade selection.

Grade refers to the severity of the AE. The CTCAE

Grade 5 (Death) is not appropriate for some AEs
displays Grades 1 through 5 with unique clinical
and therefore is not an option.

### ctivities of Daily Living (ADL)

Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the

Self care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking

<sup>†</sup> CTCAE v4.0 incorporates certain elements of the MeduRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.com).

### CONTENTS

| SOC | Page |
|---------------------------------------------------------------------|------|
| Blood and lymphatic system disorders | 3 |
| Cardiac disorders | 4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 9 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | 76 |
| Vascular disorders | 77 |

| | В | lood and lymphatic system | em disorders | | |
|---|---|---|---|---|---|
| | | | Grade | T | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| nemia | Hemoglobin (Hgb) <lln -="" 10.0="" 100="" 6.2="" <lln="" dl;="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 - 8.0 g/dL; &lt;6.2 - 4.9 mmol/L; &lt;100 - 80g/L</td><td>Hgb &lt;8.0 g/dL; &lt;4.9 mmol/L; &lt;80 g/L; transfusion indicated</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9 mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ted by an reduction in the amount of the palpitations of the heart, soft syst | • | • • • | ay include pallor of the skin and m | nucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25% reduction from normal cellularity for age | Moderately hypocellular or >25 -<br><50% reduction from normal<br>cellularity for age | Severely hypocellular or >50 -<br><=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder characteriz | ed by the inability of the bone mar | row to produce hematopoietic ele | ments. | | |
| Disseminated intravascular coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences; urgent intervention indicated | Death |
| | red by systemic pathological activa<br>s depleted of platelets and coagula | | which results in clot formation thro | oughout the body. There is an inci | ease in the |
| Febrile neutropenia | - | - | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >=38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>degrees F) for more than one ho | ed by an ANC <1000/mm3 and a sour. | single temperature of >38.3 degre | es C (101 degrees F) or a sustaine | ed temperature of >=38 degrees 0 | C (100.4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and >=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that in | ndicate widespread erythrocyte ce | Il membrane destruction. | | |
| Hemolytic uremic syndrome | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder characteriz | ed by a form of thrombotic microal | ngiopathy with renal failure, hemo | lytic anemia, and severe thromboo | cytopenia. | |
| Leukocytosis | - | - | >100,000/mm3 | Clinical manifestations of leucostasis; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by laboratory test results that ir | ndicate an increased number of w | nite blood cells in the blood. | | |
| Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in a lymph node. | | | |
| Spleen disorder | Incidental findings (e.g., Howell-<br>Jolly bodies); mild degree of<br>thrombocytosis and<br>leukocytosis | Prophylactic antibiotics indicated | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder of the splee | en. | | | | |
| Thrombotic thrombocytopenic<br>ourpura | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | - | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | ted by the presence of microangiop | • | cytopenic purpura, fever, renal abr | normalities and neurological abnor | malities suc |
| | ual disturbances. It is an acute or s | subacute condition. | Τ | Τ | 1 |
| Blood and lymphatic system<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Grade | | | | | |
|---|---|---|---|---|---|
| A d | | | I | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute coronary syndrome | | Symptomatic, progressive angina; cardiac enzymes normal; hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | zed by signs and symptoms related<br>unstable angina to myocardial infa | • | lium secondary to coronary artery | disease. The clinical presentation | covers a |
| Aortic valve disease | Asymptomatic valvular | Asymptomatic; moderate | Symptomatic; severe | Life-threatening consequences; | Death |
| | thickening with or without mild | regurgitation or stenosis by | regurgitation or stenosis by | urgent intervention indicated | |
| | valvular regurgitation or | imaging | imaging; symptoms controlled | (e.g., valve replacement, | |
| | stenosis by imaging | | with medical intervention | valvuloplasty) | |
| Definition: A disorder characteriz | zed by a defect in aortic valve func | tion or structure. | | | |
| Asystole | Periods of asystole; non-urgent | = | - | Life-threatening consequences; | Death |
| · | medical management indicated | | | urgent intervention indicated | |
| Definition: A disorder characteriz | zed by a dysrhythmia without cardi | ac electrical activity. Typically, this | is accompanied by cessation of the | he pumping function of the heart. | • |
| Atrial fibrillation | Asymptomatic, intervention not | Non-urgent medical intervention | | Life-threatening consequences; | Death |
| | indicated | indicated | controlled medically, or controlled with device (e.g., pacemaker), or ablation | urgent intervention indicated | _ 5601 |
| Definition: A disorder characteriz originates above the ventricles. | zed by a dysrhythmia without disce | ernible P waves and an irregular ve | entricular response due to multiple | reentry circuits. The rhythm distur | bance |
| Atrial flutter | Asymptomatic, intervention not | Non-urgent medical intervention | Symptomatic and incompletely | Life-threatening consequences; | Death |
| Alliai liullei | indicated | indicated | controlled medically, or | urgent intervention indicated | Dealii |
| | indicated | indicated | controlled with device (e.g., | digent intervention indicated | |
| | | | pacemaker), or ablation | | |
| Definition: A disorder characteriz | ed by a dysrhythmia with organize | ed rhythmic atrial contractions with | a rate of 200-300 beats per minut | e. The rhythm disturbance origina | tes in the |
| atria. | , , , | , | · | , | |
| Atrioventricular block complete | - | Non-urgent intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., | Life-threatening consequences; urgent intervention indicated | Death |
| | | | pacemaker) | | |
| | zed by a dysrhythmia with complete | | conduction through the AV node t | to the ventricles. | |
| Atrioventricular block first | Asymptomatic, intervention not | Non-urgent intervention | - | - | - |
| degree | indicated | indicated | | | |
| | zed by a dysrhythmia with a delay i<br>interval greater than 200 milliseco | • | tion of an electrical impulse throug | gh the atrioventricular (AV) node b | eyond 0. |
| Cardiac arrest | - | - | - | Life-threatening consequences; | Death |
| | | | | urgent intervention indicated | |
| Definition: A disorder characteriz | zed by cessation of the pumping fu | inction of the heart. | | | |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting | Pain at rest; limiting self care | - | - |
| D 6 W A W | | instrumental ADL | ADL | I | I |
| | zed by substernal discomfort due to | 1 | | I | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by pathological irregularities in | the cardiac conduction system. | | | |
| Constrictive pericarditis | - | - | Symptomatic heart failure or | Refractory heart failure or other | Death |
| | | | other cardiac symptoms, responsive to intervention | poorly controlled cardiac symptoms | |
| | | | • | | • |
| Definition: A disorder characteriz | lzed by a thickened and fibrotic peri | icardial sac; these fibrotic changes | impede normal myocardial function | on by restricting myocardial muscle | e action. |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic<br>dysfunction | - | - | Symptomatic due to drop in ejection fraction responsive to intervention | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated | Death |
| | ed by failure of the left ventricle to<br>nea, orthopnea, and other signs ar | | an increase in distending pressurestion and edema. | e and in end-diastolic volume. Clir | nical |
| Mitral valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in mitral valve funct | tion or structure. | 1 | T | |
| Mobitz (type) II atrioventricular<br>block | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with relatively atrioventricular (AV) node to the ve | | block of an atrial impulse. This is the | he result of intermittent failure of a | trial electrica |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a progre<br>on through the atrioventricular (AV | | ior to the blocking of an atrial impu | lse. This is the result of intermitter | nt failure of |
| Myocardial infarction | - | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences;<br>hemodynamically unstable | Death |
| Definition: A disorder characteriz | ed by gross necrosis of the myoca | rdium; this is due to an interruptio | on of blood supply to the area. | ' | • |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characteriz | ed by inflammation of the muscle | tissue of the heart. | | • | |
| Palpitations | Mild symptoms; intervention not indicated | Intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by an unpleasant sensation of | irregular and/or forceful beating o | f the heart. | | |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characteriz<br>originates in the atria. | ed by a dysrhythmia with abrupt o | nset and sudden termination of at | rial contractions with a rate of 150- | 250 beats per minute. The rhythm | n disturbance |
| Pericardial effusion | - | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by fluid collection within the pe | ricardial sac, usually due to inflam | mation. | | |
| Pericardial tamponade | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an increase in intrapericardi | al pressure due to the collection of | of blood or fluid in the pericardium. | Γ | T |
| Pericarditis | Asymptomatic, ECG or physical findings (e.g., rub) consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic consequences (e.g., pericardial constriction) | Life-threatening consequences; urgent intervention indicated | Death |

| | | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis by imaging; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteriz | ed by a defect in pulmonary valve | function or structure. | | _ | |
| Restrictive cardiomyopathy | | to fill with blood because the much | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other poorly controlled cardiac symptoms | Death |
| | red by an inability of the ventricles | 1 | 1 ' | · · | l <sub>n "</sub> |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., ventricular assist device);<br>heart transplant indicated | Death |
| | ed by impairment of right ventricul | ar function associated with low eje | ection fraction and a decrease in m<br>T | notility of the right ventricular wall. | |
| Sick sinus syndrome | Asymptomatic, intervention not indicated | Non-urgent intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | red by a dysrhythmia with alternation | | 1 | | I |
| Sinus bradycardia | Asymptomatic, intervention not indicated | Symptomatic, medical intervention indicated | Severe, medically significant,<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by a dysrhythmia with a heart r | i · | T T | | |
| Sinus tachycardia | Asymptomatic, intervention not indicated | Symptomatic; non-urgent medical intervention indicated | Urgent medical intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates in the sinus no | ode. | |
| Supraventricular tachycardia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates above the ven | tricles. | |
| Tricuspid valve disease | Asymptomatic valvular thickening with or without mild valvular regurgitation or stenosis | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe regurgitation or stenosis; symptoms controlled with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characterize | ed by a defect in tricuspid valve fu | nction or structure. | | 1 | |
| Ventricular arrhythmia | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by a dysrhythmia that originate | s in the ventricles. | | | |
| Ventricular fibrillation | - | - | - | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz ventricles. | ed by a dysrhythmia without disce | rnible QRS complexes due to rapi | d repetitive excitation of myocardi | al fibers without coordinated contr | action of the |
| Ventricular tachycardia | - | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates distal to the bu | undle of His. | |
| Wolff-Parkinson-White<br>syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically or controlled with procedure | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of an accesso | ry conductive pathway between th | e atria and the ventricles that caus | ses premature ventricular activation | n. |
| Cardiac disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Congenital, familial and genetic disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 2 3 4 | | | | |
| Congenital, familial and genetic | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| disorders - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| i | | | disabling; limiting self care ADL | | |

| | | Ear and labyrinth dis | sorders | | |
|---|---|---|---|---|---|
| | | · | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in the ear. | | | |
| External ear inflammation | External otitis with erythema or dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis;<br>stenosis or osteomyelitis;<br>necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation, swelling and r | edness to the outer ear and ear c | anal. | ' | • |
| External ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the external ear region. | | | |
| Hearing impaired | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: subjective change in hearing in the absence of documented hearing loss. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 8 kHz in at least one ear. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 4 kHz and above in at least one ear. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of >25 dB averaged at 3 contiguous test frequencies in at least one ear; therapeutic intervention indicated. Adults not enrolled in Monitoring Program: hearing loss with hearing aid or intervention indicated; limiting self care ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): hearing loss sufficient to indicate therapeutic intervention, including hearing | Adults: Decrease in hearing to profound bilateral loss (absolute threshold >80 dB HL at 2 kHz and above); non-servicable hearing. Pediatric: Audiologic indication for cochlear implant and additional speech-language related services indicated. | - |
| Definition: A disorder characteriz<br>Middle ear inflammation | ted by partial or complete loss of the | ne ability to detect or understand s<br>Serous otitis, medical | aids; threshold shift >20 dB at 3 kHz and above in at least one ear; additional speech-language related services indicated. ounds resulting from damage to e. Mastoiditis; necrosis of canal | Life-threatening consequences; | Death |
| | | intervention indicated | soft tissue or bone | urgent intervention indicated | |
| Tinnitus | mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| | ed by noise in the ears, such as rir | | | | |
| Vertigo | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz vertigo). | led by a sensation as if the externa | 1 | ı | I<br>he himself were revolving in space | l<br>e (subjective |
| Vestibular disorder | - | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by dizziness, imbalance, nause | ea, and vision problems. | 1 | 1 | 1 |
| Ear and labyrinth disorders -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Endocrine disord | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adrenal insufficiency | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rs when the adrenal cortex does not ison's disease or primary adrenal in: | · - | cortisol and in some cases, the ho | rmone aldosterone. It may be due | to a disorder |
| Cushingoid | Mild symptoms; intervention not indicated | | Severe symptoms, medical intervention or hospitalization indicated | - | - |
| Definition: A disorder character osteoporosis, usually due to ex | rized by signs and symptoms that re | semble Cushing's disease or synd | drome: buffalo hump obesity, striat | ions, adiposity, hypertension, diab | etes, and |
| Delayed puberty | - | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age 14 yrs for females; no increase in testes volume or no Tanner Stage 2 by age 16 yrs for males; hormone replacement indicated | - | - |
| Definition: A disorder character | rized by unusually late sexual maturi | ity. | 1 | ı | 1 |
| Growth accelerated | - | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | - | - |
| Definition: A disorder character | rized by greater growth than expecte | ed for age. | | | |
| Hyperparathyroidism | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character the blood). | rized by an increase in production of | 1 | thyroid glands. This results in hype | ।<br>ercalcemia (abnormally high levels | of calcium ir |
| Hyperthyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid suppression therapy indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by excessive levels of thyroid h | normone in the body. Common ca | uses include an overactive thyroid | gland or thyroid hormone overdos | e. |
| Hypoparathyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; medical intervention or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by a decrease in production of | parathyroid hormone by the parat | hyroid glands. | | |
| Hypothyroidism | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thyroid replacement indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by a decrease in production of | , , , | and. | | 1 |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical markers of puberty for females <8 years and males <9 years | - | - | - |
| Definition: A disorder character 9 for boys. | rized by unusually early developmer | nt of secondary sexual features; th | e onset of sexual maturation begir | ns usually before age 8 for girls an | d before age |
| Virilization | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | rized by inappropriate masculinization | on occurring in a female or prepub | ertal male. | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Bistreet Vestor Adverse Event Intervention not indicated expert Appropriate and the control of diagnostic characterized by a partial of the control of th | | | Eye dis | sorders | | |
|---|---|---|---|---|---|---|
| Intervention not indicated Symptomatic, reliniting instrumental ADL Symptomatic with marked diagnostic observations only incorporated ADL Symptomatic with marked diagnostic observations only incorporate or tuzzy images. | | | - | Grade | - | |
| Definition: A disorder characterized by visual pencegoin of invating of target or face or face of target or face or face or face of target or face or fa | Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Appropriate center of disposition for indicated intervention and indicated intervention and indicated intervention and indicated intervention and indicated intervention indicated (e.g., autoract surgery) (2040 or better) Definition: A disorder characterized by partial or complete opacity of the crystalline lens of one or both eyes. This results in a decrease in visual acuity and eventual blindness if universal intervention indicated (e.g., autoract surgery). Definition: A disorder characterized by inflammation, aveiling and eventual blindness if universal intervention indicated (e.g., intervention and indicated intervention indicated (e.g., intervention indicated) (e.g., in | | | instrumental ADL | Limiting self care ADL | - | - |
| diagnostic observations only. decrease in visual acuity doverse hara 202000; operative intervention not indicated (a publicated specification of the crystalline lens of one or both eyes. This results in a decrease in visual acuity and eventual bilindness of uniterated. Lonjunctivitis Asymptomatic or mild symptomatic or mild symptoms; intervention indicated (e.g., antibiotics) insuring lens or one or both eyes. This results in a decrease in visual acuity and eventual bilindness of uniterated and symptoms; intervention indicated (e.g., antibiotics) insuring lens or one or both eyes. This results in a decrease in visual acuity and eventual bilindness of unitervention indicated (e.g., antibiotics) insuring lens or one or both eyes. This results in a decrease in visual acuity and eventual bilindness of unitervention indicated (e.g., antibiotics) insuring lens or one or both eyes. This results in a decrease in visual acuity and eventual bilindness of the content of the eye. Definition: A disorder characterized by an area of eighthelial transvention indicated (e.g., antibiotics) insuring lens or expenditure or expendi | | | | I | | |
| Definition: A disorder characterized by partial or complete opacity of the crystalline lens of one or both eyes. This results in a decrease in visual acuity and eventual blindness if untriversition and intervention indicated (e.g., definition). A graph of the crystalline lens of one or both eyes. This results in a decrease in visual acuity and eventual blindness if untriversition indicated (e.g., definition). A graph of the crystalline lens of one or both eyes. This results in a decrease in visual acuity and eventual blindness if untriversition indicated (e.g., definition). A disorder characterized by inflammation, evening and rodness to the conjunctive of the eye. Corneal ulcer - | Cataract | diagnostic observations only; | decrease in visual acuity | decrease in visual acuity<br>(worse than 20/40 but better<br>than 20/200); operative<br>intervention indicated (e.g., | , | - |
| Conjunctivities Asymptomatic or mild included (a.g., symptomatic) indicated (a.g., special agents); limiting indicated (a.g., special agents); limiting and redness to the conjunctive of the eye. Definition: A disorder characterized by an area of epithelial issue loss on the surface of the comea. It is associated with inflammatory cells in the comea and anterior chamber. | | l<br>erized by partial or complete op | l<br>acity of the crystalline lens of c | | l<br>na decrease in visual acuity ar | I<br>nd eventual blindness if |
| Symptomatic: medical (a.g., declining vision (worse than 20/200) and the proposal parts (in limiting part (are ADL: declining vision (worse than 20/200) affected expansion (worse than 20/200) affected expansion (and the proposal agents); limiting instrumental ADL (agents) and the proposal parts (agents) and the pro | | symptoms; intervention not | intervention indicated (e.g., antibiotics); limiting | Limiting self care ADL | - | - |
| Intervention indicated (e.g., obcal appets); limiting instrumental ADL perintion: A disorder characterized by an area of epithelial its loss on the surface of the cornea, it is associated with inflammatory cells in the cornea and anterior chamber. Definition: A disorder characterized by dryness of the cornea and conjunctiva. Extraocular muscle paresis Asymptomatic, clinical or dispnostic observations only instrumental ADL perintion: A disorder characterized by incomplete paralysis of an extraocular muscle. Extraocular muscle paresis Asymptomatic, clinical or dispnostic observations only instrumental ADL perintion: A disorder characterized by incomplete paralysis of an extraocular muscle. Extraocular muscle paresis Mild pain Moderate pair, limiting M | Definition: A disorder characte | erized by inflammation, swelling | and redness to the conjunctiv | a of the eye. | | |
| Dry eye Asymptomatic; clinical or diagnostic observations only; mild symptoms relieved by lubricants Definition: A disorder characterized by dryness of the come and conjunctiva. Extraocular muscle paresis Asymptomatic; clinical or diagnostic observations only instrumental ADL Limiting self care ADL; - - - | Corneal ulcer | - | intervention indicated (e.g., topical agents); limiting | declining vision (worse than | (20/200 or worse) in the | - |
| diagnostic observations only; lubricants (capital part of the part | Definition: A disorder characte | erized by an area of epithelial ti | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the cornea | and anterior chamber. |
| Extraocular muscle paresis | Dry eye | diagnostic observations only;<br>mild symptoms relieved by | agents indicated; limiting | (<20/40); limiting self care | - | - |
| Definition: A disorder characterized by incomplete paralysis of an extraocular muscle. Eye pain Mild pain Moderate pain; limiting instrumental ADL are ADL are ADL Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention indicated; limiting instrumental ADL indicated (Indicated Indicated Ind | Definition: A disorder characte | erized by dryness of the cornea | and conjunctiva. | | | |
| Eye pain Mild pain Moderate pain; limiting instrumental ADL care ADL care ADL Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention indicated; limiting instrumental ADL limiting self care ADL; operative intervention indicated; limiting instrumental ADL limiting self care ADL Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit in ovisual field deficit (limiting instrumental ADL) Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting intrumental ADL limiting self care ADL Symptomatic; medical intervention indicated; limiting self care ADL Symptomatic; medical intervention of the aqueous humor outflow. Elevated intraocular pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents; limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Extraocular muscle paresis | | • • | | - | - |
| Definition: A disorder characterized by a sensation of marked discomfort in the eye. Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated (limiting instrumental ADL) Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by a nindividual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit no visual field deficit EIOP causing early visual field spots and intervention indicated; limiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic; dinical or dispersion of marked discomfort in the eye. Night blindness Symptomatic but not limiting linitrumental ADL Limiting self care ADL Limiting self care ADL | Definition: A disorder characte | erized by incomplete paralysis of | of an extraocular muscle. | Г | I | |
| Eyelid function disorder Asymptomatic; clinical or diagnostic observations only; intervention not indicated intervention not indicated intervention indicated; limiting instrumental ADL Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit; multiple topical or oral agents indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting ADL Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit; multiple topical intervention indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting Instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Instrumental ADL Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL Decine in vision (worse than 20/40 but better than 20/2000); limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Instrumental ADL Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Eye pain | Mild pain | | | - | - |
| diagnostic observations only, intervention not indicated; limiting instrumental ADL Definition: A disorder characterized by impaired eyelid function. Flashing lights Symptomatic but not limiting ADL Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Glaucoma Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit individual seeing or or al agents indicated; limiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic but not limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Limiting self care ADL | Definition: A disorder characte | erized by a sensation of marked | d discomfort in the eye. | T | <u> </u> | 1 |
| Flashing lights | Eyelid function disorder | diagnostic observations only; | intervention indicated; | operative intervention | - | - |
| Definition: A disorder characterized by a sudden or brief burst of light. Floaters Symptomatic but not limiting ADL Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit Imiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis Symptomatic: medical intervention indicated (e.g., topical agents): limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Limiting self care ADL Limiting self care ADL | | | | I | | 1 |
| Symptomatic but not limiting ADL | Flashing lights | | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder characterized by an individual seeing spots before their eyes. The spots are shadows of opaque cell fragments in the vitreous humor or lens. Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficit no visual field deficit Fertilition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. EIOP causing early visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Keratitis - Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | | | | T | | T |
| Elevated intraocular pressure (EIOP) with single topical agent for intervention; no visual field deficits (multiple topical limiting instrumental ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents indicated (e.g., topical agents); limiting instrumental ADL EIOP causing marked visual field deficits (e.g., involving both superior and inferior visual fields); operative intervention indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Floaters | | Limiting instrumental ADL | Limiting self care ADL | - | - |
| pressure (EIOP) with single topical agent for intervention; no visual field deficit witing instrumental ADL with a field deficit (limiting instrumental ADL with a field deficit) or oral agents indicated; limiting self care ADL Definition: A disorder characterized by an increase in pressure in the eyeball due to obstruction of the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents in the aqueous humor outflow. Symptomatic; medical intervention indicated (e.g., topical agents); limiting agents in the aqueous humor outflow. Decline in vision (worse than 20/40 but better than 20/200); limiting self care ADL Definition: A disorder characterized by inflammation to the cornea of the eye. Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | Definition: A disorder characte | erized by an individual seeing s | pots before their eyes. The spo | ots are shadows of opaque cell | fragments in the vitreous hum | or or lens. |
| Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL Decline in vision (worse than 20/200 or worse) in the affected eye Decline in vision (worse than 20/200 or worse) in the affected eye Decline in vision (worse than 20/200 or worse) in the affected eye Decline in vision (worse than 20/200 or worse) in the affected eye Decline in vision (worse than 20/200 or worse) in the affected eye Decline in vision (worse than 20/200 or worse) Decline in vision (worse than 20/20 | Glaucoma | pressure (EIOP) with single topical agent for intervention; | field deficits; multiple topical or oral agents indicated; | field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated; | · ' | - |
| intervention indicated (e.g., topical agents); limiting instrumental ADL 20/200); limiting self care 20/200); limiting self care ADL 20/200 or worse) in the affected eye 20/200; limiting self care ADL 20/200; l | Definition: A disorder characte | erized by an increase in pressu | re in the eyeball due to obstruc | tion of the aqueous humor out | low. | |
| Night blindness Symptomatic but not limiting Limiting instrumental ADL Limiting self care ADL Blindness (20/200 or worse) - | | - | intervention indicated (e.g.,<br>topical agents); limiting<br>instrumental ADL | 20/40 but better than 20/200); limiting self care | (20/200 or worse) in the | - |
| | Definition: A disorder characte | | ornea of the eye. | Г | | |
| | Night blindness | | Limiting instrumental ADL | Limiting self care ADL | , | - |

| | | Eye dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or diagnostic observations only | Limiting vision of the affected eye (20/40 or better) | eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| | erized by involvement of the op | 1 | ĺ | | 1 |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by swelling around the o | ptic disc.<br>T | <u> </u> | I | |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | - |
| Definition: A disorder charact | erized by fear and avoidance of | f light. | | | |
| Retinal detachment | Asymptomatic | Exudative and visual acuity 20/40 or better | Rhegmatogenous or<br>exudative detachment;<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by the separation of the | inner retina layers from the und | lerlying pigment epithelium. | | |
| Retinal tear | - | Laser therapy or pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by a small laceration of t | he retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | s and floaters. |
| Retinal vascular disorder | - | Topical medication indicated | Intravitreal medication; operative intervention indicated | - | - |
| Definition: A disorder charact | erized by pathological retinal bl | ood vessels that adversely affe | cts vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked<br>decrease in visual acuity<br>(worse than 20/40);<br>disabling; limiting self care<br>ADL | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder involvin | g the retina. | | | | |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better) | Symptomatic, limiting self care ADL; marked decrease in visual acuity (worse than 20/40) | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by involvement of the sc | lera of the eye. | T | T | 1 |
| Uveitis | Asymptomatic; clinical or diagnostic observations only | • | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by inflammation to the uv | vea of the eye. | Ι | Ι | T. |
| Vitreous hemorrhage | Asymptomatic or mild symptoms; clinical or diagnostic observations only | Symptomatic; limiting instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder charact | erized by blood extravasation in | nto the vitreous humor. | T | T | T |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | - | - |
| Definition: A disorder of excess | ssive tearing in the eyes; it can | be caused by overproduction of | of tears or impaired drainage of | the tear duct. | |
| Eye disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Sight-threatening<br>consequences; urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe discomfort; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by swelling of the abdomen. | | | | 1 |
| Abdominal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the abdominal region. | r | Г | 1 |
| Anal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the opening in the anal | canal to the perianal skin. | | |
| Anal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the anal region | on. | | | 1 |
| Anal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the mucous | membrane of the anus. | T | <u> </u> | 1 |
| Anal necrosis | - | a in the engl region | TPN or hospitalization indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by a necrotic process occurring | | Sovere pain: limiting colf care | | |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | erized by a sensation of marked disco | | 0 , , , , | Let up a control of the control of t | Б. " |
| Anal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated; TPN or hospitalization<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the anal canal. | | | |
| Anal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ory and necrotic erosive lesion on t | he mucosal surface of the anal ca | nal. | |
| Ascites | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; invasive intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by accumulation of serous or h | emorrhagic fluid in the peritoneal | cavity. | • | • |
| Bloating | No change in bowel function or oral intake | Symptomatic, decreased oral intake; change in bowel function | - | - | - |
| Definition: A disorder characte | rized by subject-reported feeling of ι | ncomfortable fullness of the abdo | men. | • | • |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the cecum. | | | • | • |
| Cheilitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | - | - |
| | | 1 | I . | ı | I |

| Gastrointestinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| Advance France | | | | | Ι, |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Colitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the colon. | | | | |
| Colonic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the large intestine and | another organ or anatomic site. | | |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the colon. | T | T | Г | |
| Colonic obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated rized by blockage of the normal flow | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | Tized by blockage of the normal flow | | | | D41- |
| Colonic perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by a rupture in the colonic wall. | | | | |
| Colonic stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the colon. | ' | ' | • |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the colon. | | |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with regular use of laxatives or enemas; limiting instrumental ADL | Obstipation with manual evacuation indicated; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by irregular and infrequent or d | ifficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis or periapical abscess or resulting in tooth loss | - | - |
| Definition: A disorder characte | rized by the decay of a tooth, in whice | h it becomes softened, discolored | and/or porous. | | |
| Diarrhea | Increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day over baseline; moderate increase in ostomy output compared to baseline | Increase of >=7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by frequent and watery bowel r | novements. | | | |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dietary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment orally; tube feeding or TPN indicated; unstimulated saliva <0.1 ml/min | - | - |

| | Gastrointestinal disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the duodenum and and | ther organ or anatomic site. | | |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by bleeding from the duodenur | | 1 | | |
| Duodenal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective operative intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by blockage of the normal flow | of stomach contents through the | duodenum. | | |
| Duodenal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a rupture in the duodenal w | all. | - | 1 | 1 |
| Duodenal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the duodenum. | | | |
| Duodenal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a circumscribed, inflammato | l e | | nal wall. | 1 |
| Dyspepsia | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| Definition: A disorder characte<br>neartburn, nausea and vomitir | rized by an uncomfortable, often pai | nful feeling in the stomach, resulti | ng from impaired digestion. Sympt | oms include burning stomach, blo | ating, |
| Dysphagia | Symptomatic, able to eat regular diet | Symptomatic and altered eating/swallowing | Severely altered eating/swallowing; tube feeding or TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by difficulty in swallowing. | | | | |
| Enterocolitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Abdominal pain; mucus or blood in stool | Severe or persistent abdominal pain; fever; ileus; peritoneal signs | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation of the small ar | nd large intestines. | | 1 | |
| Enterovesical fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | n between the urinary bladder and | the intestine. | | |
| Esophageal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | n between the esophagus and and | other organ or anatomic site. | | |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | · · | • | • | • | • |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a necrotic process occurring | g in the esophageal wall. | | | |
| Esophageal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by blockage of the normal flow | of the contents in the esophagus | i.<br>T | T | |
| Esophageal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the esophageal region. | | | |
| Esophageal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a rupture in the wall of the e | 1 | 1 | <u> </u> | |
| Esophageal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the esophagus. | | | |
| Esophageal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the esopha | geal wall. | |
| Esophageal varices<br>hemorrhage | - | Self-limited; intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from esophageal v | rarices. | | | |
| Esophagitis Definition: A disorder character | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered eating/swallowing; oral supplements indicated | Severely altered<br>eating/swallowing; tube feeding,<br>TPN or hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Fecal incontinence | Occasional use of pads required | | Severe symptoms; elective | - | - |
| | | | operative intervention indicated | | |
| Definition: A disorder characte | rized by inability to control the escap | e of stool from the rectum. | T | T | |
| Flatulence | Mild symptoms; intervention not indicated | Moderate; persistent; psychosocial sequelae | - | - | - |
| Definition: A disorder characte | rized by a state of excessive gas in | the alimentary canal. | | | |
| Gastric fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>bowel rest; tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | n between the stomach and anoth | ner organ or anatomic site. | T | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the gastric wa | all. | | | |
| Gastric necrosis | - | - | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | 1 | • | • | 1 | |

| | Gastrointestinal disorders | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation Definition: A disorder character | rized by a rupture in the stomach wa | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | | | Soverely altered Cl function: | Life threatening concequences: | Death |
| Gastric stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Deam |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the stomach. | | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; medical intervention<br>indicated; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by a circumscribed, inflammato | T | the mucosal surface of the stomac | | 1 |
| Gastritis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by inflammation of the stomach | ).<br>! | 1 | I | |
| Gastroesophageal reflux<br>disease | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms; surgical intervention indicated | - | - |
| | rized by reflux of the gastric and/or d<br>y result in injury to the esophageal m | | | nd usually caused by incompetend | e of the lo |
| Gastrointestinal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site. | |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the gastrointestinal region | 1. | | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to maintain nutrition with dietary and lifestyle modifications; may need pharmacologic intervention | Weight loss; refractory to medical intervention; unable to maintain nutrition orally | - | - |
| Definition: A disorder characte | rized by an incomplete paralysis of the | he muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small into | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with oral intake | Severe pain; inability to aliment orally | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in the gingival region. | T | T | |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the hemorrho | ids. | | | |
| Hemorrhoids | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characte | rized by the presence of dilated vein | s in the rectum and surrounding a | rea. | | |
| leal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the ileum and another o | organ or anatomic site. | | |
| leal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical | Transfusion, radiologic, | Life-threatening consequences; | Death |
| Ç | | intervention or minor cauterization indicated | endoscopic, or elective operative intervention indicated | urgent intervention indicated | |

| Gastrointestinal disorders Grade | | | | | |
|---|---|---|---|---|---|
| | | | | | Τ. |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| leal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents in the ile | eum. | | |
| lleal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a rupture in the ileal wall. | | | | |
| lleal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a narrowing of the lumen of | the ileum. | | Т | |
| lleal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the ileum. | <u> </u> | |
| lleus<br>Definition: A disorder characteri: | -<br>zed by failure of the ileum to transp | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Intra-abdominal hemorrhage | - | Medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ा<br>zed by bleeding in the abdominal c | avity. | 1. | ı | ' |
| Jejunal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ा<br>zed by an abnormal communicatio। | ।<br>n between the jejunum and anoth | 1 | ı | 1 |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | zed by bleeding from the jejunal wa | il. | | ' | • |
| Jejunal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered Gl function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by blockage of the normal flow | of the intestinal contents in the je | ejunum. | | |
| Jejunal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ਾ<br>zed by a rupture in the jejunal wall. | · | <u> </u> | ·<br> | |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a narrowing of the lumen of | the jejunum. | | | |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | zed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the jejunun | n. | · |
| Lip pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Lower gastrointestinal<br>hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the lower gas | strointestinal tract (small intestine, | large intestine, and anus). | | • |
| Malabsorption | - | Altered diet; oral intervention indicated | Inability to aliment adequately;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inadequate absorption of nu | trients in the small intestine. Sym | ptoms include abdominal marked | discomfort, bloating and diarrhea. | |
| Mucositis oral | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Moderate pain; not interfering with oral intake; modified diet indicated | Severe pain; interfering with oral intake | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the oral mu | cosal. | | | 1 |
| Nausea | Loss of appetite without alteration in eating habits | Oral intake decreased without significant weight loss, dehydration or malnutrition | Inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated | - | - |
| Definition: A disorder characte | erized by a queasy sensation and/or | the urge to vomit. | T | T | |
| Obstruction gastric | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of the contents in the stomach. | | | |
| Oral cavity fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | between the oral cavity and ano | ther organ or anatomic site. | | |
| Oral dysesthesia | Mild discomfort; not interfering with oral intake | Moderate pain; interfering with oral intake | Disabling pain; tube feeding or TPN indicated | - | - |
| | erized by a burning or tingling sensati | on on the lips, tongue or entire mo | outh. | Ī | 1 |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the mouth. | | | | |
| Oral pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the mouth, tongue or lips | | | |
| Pancreatic duct stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | rized by a narrowing of the lumen of | the pancreatic duct. | | | |
| Pancreatic fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by an abnormal communication | | 1 | | 1 |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the pancreas | T | _ | T | |
| Pancreatic necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a necrotic process occurring | g in the pancreas. | _ | _ | |
| Pancreatitis | - | Enzyme elevation or radiologic findings only | Severe pain; vomiting; medical intervention indicated (e.g., analgesia, nutritional support) | Life-threatening consequences; urgent intervention indicated | Death |

| | | Gastrointestinal dis | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte | erized by inflammation of the pancrea | S. | 1 | | |
| Periodontal disease | Gingival recession or gingivitis;<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or<br>gingivitis; multiple sites of<br>bleeding on probing; moderate<br>bone loss | Spontaneous bleeding; severe bone loss with or without tooth loss; osteonecrosis of maxilla or mandible | - | - |
| Definition: A disorder in the gi | ngival tissue around the teeth. | | | | |
| Peritoneal necrosis | - | - | Tube feeding or TPN indicated; radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a necrotic process occurring | in the peritoneum. | | | |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the rectum. | | | | |
| Rectal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the rectum and anothe | r organ or anatomic site. | | |
| Rectal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the rectal wal | and discharged from the anus. | 1 | <u> </u> | |
| Rectal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |
| | erized by inflammation of the mucous | membrane of the rectum. | | | |
| Rectal necrosis | - | - | Tube feeding or TPN indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of the intestinal contents in the re | ctum. | Г | |
| Rectal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| | erized by a sensation of marked disco | | 1_ | | _ |
| Rectal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a rupture in the rectal wall. | | T. | <b>,</b> | |
| Rectal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the rectum. | | | |
| Rectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function (e.g. altered dietary habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Retroperitoneal hemorrhage | -<br>led by bleeding from the retroperite | Self-limited; intervention indicated | Transfusion, medical, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | T . | | Acute colivery aland necresis. | Life threatening concessions | Dooth |
| Salivary duct inflammation | Slightly thickened saliva; slightly altered taste (e.g., metallic) | Thick, ropy, sticky saliva;<br>markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis;<br>severe secretion-induced<br>symptoms (e.g., thick saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated;<br>limiting self care ADL; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the salivary | duct. | 1 | | |
| Salivary gland fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal mucositis | Asymptomatic or mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe pain; interfering with oral<br>intake; tube feeding, TPN or<br>hospitalization indicated; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the normal flow | of the intestinal contents. | | | |
| Small intestinal perforation | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the small intesti | ne wall. | | | |
| Small intestinal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the lumen of | the small intestine. | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the small in | ntestine. | |
| Stomach pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the stomach. | 1 | r | |
| Tooth development disorder | Asymptomatic; hypoplasia of tooth or enamel | Impairment correctable with oral surgery | Maldevelopment with impairment not surgically correctable; disabling | - | - |
| Definition: A disorder characteriz | ed by a pathological process of the | e teeth occurring during tooth dev | elopment. | I | 1 |
| Tooth discoloration | Surface stains | - | - | - | - |
| Definition: A disorder characteriz | ed by a change in tooth hue or tint | t. | 1 | 1 | |
| Toothache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care | - | - |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Typhlitis | - | - | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal signs | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation of the cecum. | | | | |
| Upper gastrointestinal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical intervention or minor cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the upper gas | trointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | |
| Vomiting | 1 - 2 episodes (separated by 5 minutes) in 24 hrs | 3 - 5 episodes (separated by 5 minutes) in 24 hrs | >=6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the reflexive act of ejecting t | he contents of the stomach throug | gh the mouth. | • | |
| Gastrointestinal disorders -<br>Other, specify | , , , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold; | Moderate tremor of the entire | Severe or prolonged, not | | |
| O.I.I.I.G | shivering; chattering of teeth | body; narcotics indicated | responsive to narcotics | | |
| Definition: A disorder characte | erized by a sensation of cold that ofte | n marks a physiologic response to | sweating after a fever. | | • |
| Death neonatal | = | = | = | - | Death |
| Definition: A disorder characte | erized by cessation of life occurring d | uring the first 28 days of life. | ' | ' | |
| Death NOS | - | - | - | - | Death |
| Definition: A cessation of life | that cannot be attributed to a CTCAE | term associated with Grade 5. | ' | ' | , |
| Edema face | Localized facial edema | Moderate localized facial | Severe swelling; limiting self | - | - |
| | | edema; limiting instrumental | care ADL | | |
| | | ADL | | | |
| Definition: A disorder characte | erized by swelling due to excessive flu | uid accumulation in facial tissues. | 1 | T | |
| Edema limbs | 5 - 10% inter-limb discrepancy | >10 - 30% inter-limb | >30% inter-limb discrepancy in | - | - |
| | in volume or circumference at | discrepancy in volume or | volume; gross deviation from | | |
| | point of greatest visible difference; swelling or | circumference at point of greatest visible difference; | normal anatomic contour;<br>limiting self care ADL | | |
| | obscuration of anatomic | readily apparent obscuration of | | | |
| | architecture on close inspection | anatomic architecture; | | | |
| | | obliteration of skin folds; readily | | | |
| | | apparent deviation from normal | | | |
| | | anatomic contour; limiting | | | |
| | | instrumental ADL | | | 1 |
| | erized by swelling due to excessive flo | 1 | | | 1 |
| Edema trunk | Swelling or obscuration of | Readily apparent obscuration of | Gross deviation from normal | - | - |
| | anatomic architecture on close inspection | anatomic architecture;<br>obliteration of skin folds; readily | anatomic contour; limiting self care ADL | | |
| | Парссион | apparent deviation from normal | Carc ADL | | |
| | | anatomic contour; limiting | | | |
| | | instrumental ADL | | | |
| Definition: A disorder characte | erized by swelling due to excessive flo | uid accumulation in the trunk area. | | | |
| Facial pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | - |
| | | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by a sensation of marked disco | omfort in the face. | | | |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest; | Fatigue not relieved by rest, | - | - |
| | | limiting instrumental ADL | limiting self care ADL | | |
| Definition: A disorder characte | erized by a state of generalized weak | ness with a propounced inability to | summon sufficient energy to acc | omplish daily activities. | |
| | enzed by a state of generalized weak | ricss with a profited feed mability to | | | |
| | | >39.0 - 40.0 degrees C (102.3 - | >40.0 degrees C (>104.0 | >40.0 degrees C (>104.0 | Death |
| | | | | >40.0 degrees C (>104.0 degrees F) for >24 hrs | Death |
| Fever | 38.0 - 39.0 degrees C (100.4 - | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) | >40.0 degrees C (>104.0 degrees F) for <=24 hrs | , | Death |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) erature above the upper limit of not moderate symptoms; limiting | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self | , | Death - |
| Fever<br>Definition: A disorder charact | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temp | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of new control of the control o | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. | , | Death<br>- |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temp | >39.0 - 40.0 degrees C (102.3 -<br>104.0 degrees F)<br>perature above the upper limit of no<br>Moderate symptoms; limiting<br>instrumental ADL | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of no Moderate symptoms; limiting instrumental ADL r to those observed in patients with | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., wide- | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not move a support of the su | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not moderate symptoms; limiting instrumental ADL r to those observed in patients with Moderate change in gait (e.g., wide-based, limping or | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., wide- | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not moderate symptoms; limiting instrumental ADL r to those observed in patients with Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., wide- | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not moderate symptoms; limiting instrumental ADL r to those observed in patients with Moderate change in gait (e.g., wide-based, limping or | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. Gait disturbance | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., widebased, limping or hobbling) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not be a considered and the symptoms; limiting instrumental ADL To those observed in patients with the symptoms in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., widebased, limping or hobbling) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not be a considered and the symptoms; limiting instrumental ADL To those observed in patients with the symptoms in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b | degrees F) for >24 hrs | - |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. Gait disturbance Definition: A disorder character | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., widebased, limping or hobbling) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not be a support of the supp | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b Disabling; limiting self care ADL | degrees F) for >24 hrs - ody aches, malaise, loss of appeti | - ite and dr |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. Gait disturbance Definition: A disorder character | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., widebased, limping or hobbling) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not be a considered and the symptoms; limiting instrumental ADL Moderate symptoms; limiting instrumental ADL Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL 35 - >32 degrees C; 95 - >89.6 | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b Disabling; limiting self care ADL | degrees F) for >24 hrs - ody aches, malaise, loss of appeti - <=28 degrees C; 82.4 degrees | - ite and dr |
| Fever Definition: A disorder character Flu like symptoms Definition: A disorder character cough. Gait disturbance Definition: A disorder character | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) erized by elevation of the body's temporal Mild flu-like symptoms present erized by a group of symptoms simila Mild change in gait (e.g., widebased, limping or hobbling) | >39.0 - 40.0 degrees C (102.3 - 104.0 degrees F) perature above the upper limit of not be a considered and the symptoms; limiting instrumental ADL Moderate symptoms; limiting instrumental ADL Moderate change in gait (e.g., wide-based, limping or hobbling); assistive device indicated; limiting instrumental ADL 35 - >32 degrees C; 95 - >89.6 | >40.0 degrees C (>104.0 degrees F) for <=24 hrs ormal. Severe symptoms; limiting self care ADL h the flu. It includes fever, chills, b Disabling; limiting self care ADL | degrees F) for >24 hrs - ody aches, malaise, loss of appeti - <=28 degrees C; 82.4 degrees F; life-threatening | - ite and dr |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| nfusion related reaction | Mild transient reaction; infusion | Therapy or infusion interruption | Prolonged (e.g., not rapidly | Life-threatening consequences; | Death |
| illiusion relateu reaction | interruption not indicated; | indicated but responds promptly | responsive to symptomatic | urgent intervention indicated | Dealii |
| | intervention not indicated | to symptomatic treatment (e.g., | medication and/or brief | argoni intervention indicated | |
| | intervention net maieuteu | antihistamines, NSAIDS, | interruption of infusion); | | |
| | | narcotics, IV fluids); prophylactic | | | |
| | | medications indicated for <=24 | following initial improvement; | | |
| | | hrs | hospitalization indicated for | | |
| | | | clinical sequelae | | |
| Definition: A disorder characteriz | ा<br>zed by adverse reaction to the infus | ।<br>sion of pharmacological or biologic | | I | 1 |
| nfusion site extravasation | , | Erythema with associated | Ulceration or necrosis; severe | Life-threatening consequences; | Death |
| The same that are same to the | | symptoms (e.g., edema, pain, | tissue damage; operative | urgent intervention indicated | Dou |
| | | induration, phlebitis) | intervention indicated | angent intervention introduce | |
| Definition: A disorder characteriz | ।<br>zed by leakage of a pharmacologic | , | ' | I<br>ssue. Signs and symptoms include | l<br>e induratio |
| | sation and marked discomfort at the | • | madion die me and dandang a | oud. Digno una dymptomo moida | o induratio |
| njection site reaction | Tenderness with or without | Pain; lipodystrophy; edema; | Ulceration or necrosis; severe | Life-threatening consequences; | Death |
| | associated symptoms (e.g., | phlebitis | tissue damage; operative | urgent intervention indicated | |
| | warmth, erythema, itching) | | intervention indicated | | |
| Definition: A disorder characterize | zed by an intense adverse reaction | (usually immunologic) developing | ' | • | • |
| rritability | Mild; easily consolable | Moderate; limiting instrumental | Severe abnormal or excessive | - | _ |
| | inima, eachy consciusio | ADL; increased attention | response; limiting self care ADL; | | |
| | | indicated | inconsolable | | |
| Definition: A diserder characteris | ।<br>zed by an abnormal responsivenes: | ļ | 1 | l<br>ht a drug an amational situation | <br> |
| condition. | zed by an abnormal responsivenes: | s to stillfull of physiological arous | ii, may be in response to pain, mg | ni, a drug, an emotional situation ( | or a medic |
| _ocalized edema | Localized to dependent areas, | Moderate localized edema and | Severe localized edema and | - | _ |
| | no disability or functional | intervention indicated; limiting | intervention indicated; limiting | | |
| | impairment | instrumental ADL | self care ADL | | |
| Definition: A disorder characteria | 1 ' | ı | 1 | ļ | 1 |
| Delimition. A disorder characteriz | zed by swelling due to excessive flu | | offic site. | | |
| Moloico | | | | | |
| Malaise | Uneasiness or lack of well being | | | | |
| | | being; limiting instrumental ADL | faeling | | |
| Definition: A disorder characteriz | Uneasiness or lack of well being zed by a feeling of general discomfe | being; limiting instrumental ADL | | Life threatening concerns | Dooth |
| Definition: A disorder characteriz | | being; limiting instrumental ADL | Shock with azotemia and acid- | Life-threatening consequences | Death |
| Definition: A disorder characteriz | | being; limiting instrumental ADL | Shock with azotemia and acid-<br>base disturbances; significant | (e.g., vasopressor dependent | Death |
| Definition: A disorder characteriz | | being; limiting instrumental ADL | Shock with azotemia and acid- | (e.g., vasopressor dependent and oliguric or anuric or | Death |
| Definition: A disorder characteriz | | being; limiting instrumental ADL | Shock with azotemia and acid-<br>base disturbances; significant | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characteriz<br>Multi-organ failure | zed by a feeling of general discomfo | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts - | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | (e.g., vasopressor dependent and oliguric or anuric or | Death |
| Definition: A disorder characteriz<br>Multi-organ failure<br>Definition: A disorder characteriz | zed by a feeling of general discomfo | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts - the lungs, liver, kidney and clotting | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Multi-organ failure | zed by a feeling of general discomform. - zed by progressive deterioration of Asymptomatic localized neck | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities<br>g mechanisms. | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characteriz<br>Multi-organ failure<br>Definition: A disorder characteriz | zed by a feeling of general discomfo | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck); | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characteriz<br>Multi-organ failure<br>Definition: A disorder characteriz | zed by a feeling of general discomform. - zed by progressive deterioration of Asymptomatic localized neck | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities<br>g mechanisms. | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characteriz<br>Multi-organ failure<br>Definition: A disorder characteriz<br>Neck edema | zed by a feeling of general discomform. - zed by progressive deterioration of Asymptomatic localized neck edema | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities<br>g mechanisms.<br>Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize | zed by a feeling of general discomform. zed by progressive deterioration of Asymptomatic localized neck edema | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL atton of excessive fluid in the neck | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize | zed by a feeling of general discomform. - zed by progressive deterioration of Asymptomatic localized neck edema | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain | zed by a feeling of general discomformation of a symptomatic localized neck edema eled by swelling due to an accumula Mild pain | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL stion of excessive fluid in the neck Moderate pain; limiting instrumental ADL | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death - |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Definition: A disorder characterize | zed by a feeling of general discomformal dis | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL atton of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death - |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Definition: A disorder characterize | zed by a feeling of general discomformation of a symptomatic localized neck edema eled by swelling due to an accumula Mild pain | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL atton of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death - |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain | zed by a feeling of general discomformation of a symptomatic localized neck edema will be swelling due to an accumulated by swelling due to an accumulated by discomfort in the chest unrelegation. | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death - |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Pain Definition: A disorder characterize | zed by a feeling of general discomformal dis | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care<br>ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic acidosis) - | - |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Sudden death NOS | zed by a feeling of general discomformation of dealing and progressive deterioration of dealing and progressive deterioration of dealing dealing dealing due to an accumulated by swelling due to an accumulated by discomfort in the chest unreaded by discomfort in the chest unreaded by the sensation of marked discontinuous dealing deal | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care<br>ADL Severe pain; limiting self care | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Sudden death NOS Definition: An unexpected cessa | ted by a feeling of general discomformation of life that cannot be attributed. | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clotting Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. to a CTCAE term associated with | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities g mechanisms. Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL Severe pain; limiting self care<br>ADL Severe pain; limiting self care<br>ADL | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic acidosis) - | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Sudden death NOS Definition: An unexpected cessa General disorders and | zed by a feeling of general discomform. zed by progressive deterioration of Asymptomatic localized neck edema zed by swelling due to an accumulated by discomfort in the chest unreleased by the sensation of marked discomfort in the chest unrelease | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. to a CTCAE term associated with | Shock with azotemia and acid- base disturbances; significant coagulation abnormalities g mechanisms. Generalized neck edema (e.g., difficulty in turning neck); limiting self care ADL Severe pain; limiting self care ADL Severe pain; limiting self care ADL - a Grade 5. Severe or medically significant | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic acidosis) - - Life-threatening consequences; | - |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Sudden death NOS Definition: An unexpected cessa General disorders and administration site conditions - | zed by a feeling of general discomform. zed by progressive deterioration of Asymptomatic localized neck edema zed by swelling due to an accumulated by discomfort in the chest unreleff Mild pain to the chest unreleff wild pain to the chest unreleff by the sensation of marked discomposition of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention | Shock with azotemia and acid- base disturbances; significant coagulation abnormalities g mechanisms. Generalized neck edema (e.g., difficulty in turning neck); limiting self care ADL Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately life- | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic acidosis) - | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Sudden death NOS | ted by a feeling of general discomformal composition of the desired by progressive deterioration of the desired by swelling due to an accumulate discomformal composition of the desired by discomfort in the chest unrelevable discomformal composition of life that cannot be attributed asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. - to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention indicated; limiting age- | Shock with azotemia and acid- base disturbances; significant coagulation abnormalities g mechanisms. Generalized neck edema (e.g., difficulty in turning neck); limiting self care ADL Severe pain; limiting self care ADL Severe pain; limiting self care ADL - a Grade 5. Severe or medically significant but not immediately life- threatening; hospitalization or | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic acidosis) - - Life-threatening consequences; | Death |
| Definition: A disorder characterize Multi-organ failure Definition: A disorder characterize Neck edema Definition: A disorder characterize Non-cardiac chest pain Definition: A disorder characterize Pain Definition: A disorder characterize Sudden death NOS Definition: An unexpected cessa General disorders and administration site conditions - | zed by a feeling of general discomform. zed by progressive deterioration of Asymptomatic localized neck edema zed by swelling due to an accumulated by discomfort in the chest unreleff Mild pain to the chest unreleff wild pain to the chest unreleff by the sensation of marked discomposition of life that cannot be attributed Asymptomatic or mild symptoms; clinical or diagnostic | being; limiting instrumental ADL ort or uneasiness, an out-of-sorts the lungs, liver, kidney and clottin Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL ation of excessive fluid in the neck Moderate pain; limiting instrumental ADL lated to a heart disorder. Moderate pain; limiting instrumental ADL comfort, distress or agony. to a CTCAE term associated with Moderate; minimal, local or noninvasive intervention | Shock with azotemia and acid- base disturbances; significant coagulation abnormalities g mechanisms. Generalized neck edema (e.g., difficulty in turning neck); limiting self care ADL Severe pain; limiting self care ADL Severe pain; limiting self care ADL - Grade 5. Severe or medically significant but not immediately life- | (e.g., vasopressor dependent and oliguric or anuric or ischemic colitis or lactic acidosis) - - Life-threatening consequences; | Death |

| disgnostic observations only, intervention on Indicated visa from the Indicated visa superior operative intervention indicated visa superior operative intervention indicated visa superior operative intervention indicated visa | | | Hepatobiliary diso | | | |
|---|---|---|---|---|---|---|
| Bille duct stenosis a Apyropromitic citiese or disponsite contending on the formation of the field of the fie | | | | 1 | I | 1 |
| diagnosatic observations only. Introduction. If failable indicated <24 inadicated; and indicated <24 inadicated; and indicated <25 inadicated. Definition. A clasorier characterized by a narrowing of the lumen of the bile dict. Simptomatic and intervention not indicated. Simptomatic and intervention not reducted by a narrowing of the lumen of the bile dict. Simptomatic and intervention not reducted by an abnormal communication between the bile ducts and another origin or anatomic site. Cholecystitis | | | | | | |
| Symptomatic and intervention Symptomatic and intervention Symptomatic and intervention Symptomatic Sympt | Bile duct stenosis | diagnostic observations only; | function; IV fluids indicated <24 | radiologic, endoscopic or elective operative intervention | urgent operative intervention | Death |
| Definition: A disorder characterized by an abnormal communication between the bile ducts and another organ or anatomic atte. Cholecystiss - Symptomatic, medical intervention indicated of medical intervention indicated intervent | Definition: A disorder character | rized by a narrowing of the lumen of | the bile duct. | _ | | |
| Intervention indicated Intervention indica | Biliary fistula | - | 1 1 1 | TPN indicated; endoscopic intervention indicated; elective | urgent operative intervention | Death |
| Intervention indicated Intervention indica | Definition: A disorder character | rized by an abnormal communication | n between the bile ducts and anot | ner organ or anatomic site. | | |
| Salbladder fistula Asymptomatic clinical or diagnostic observations only; intervention not indicated Intervention not indicated Definition: A disorder characterized by an abnormal communication between the galibladder and another organ or anatomic site. Galibladder necrosis Life-threatening consequences; Use the contents of the galibladder and another organ or anatomic site. Galibladder obstruction Asymptomatic; clinical or diagnostic observations only; intervention indicated under the galibladder. Galibladder obstruction Asymptomatic; clinical or diagnostic observations only; intervention not indicated which is the contents of the galibladder. Galibladder pain Mild pain Mild pain Moderate pain; limiting self care Adisorder characterized by a sensation of marked discomfort in the galibladder region. Galibladder perforation Asterixis; mild encephalopathy; coma; life-threatening consequences; urgent operative intervention indicated on the galibladder region. Galibladder perforation Asterixis; mild encephalopathy; coma; life-threatening consequences; urgent intervention indicated of surfacion; by a sensation of marked discomfort in the galibladder. Galibladder perforation Asterixis; mild encephalopathy; coma; life-threatening consequences; urgent intervention indicated of surfacion; provided intervent | Cholecystitis | - | | endoscopic or elective operative | urgent operative intervention | Death |
| diagnostic observations only, intervention not indicated Gf function; TPN indicated; radiologic, endoscopic or elective operative intervention indicated urgent intervention indicated urgent intervention indicated | Definition: A disorder character | rized by inflammation involving the g | ı<br>gallbladder. It may be associated v | vith the presence of gallstones. | 1 | |
| Galibladder necrosis | Gallbladder fistula | diagnostic observations only; | 1 ' | GI function; TPN indicated; radiologic, endoscopic or elective operative intervention | urgent operative intervention | Death |
| Definition: A disorder characterized by a necrotic process occurring in the gallbladder. Gallbladder obstruction Asymptomatic; clinical or diagnostic observations only; intervention not indicated Asymptomatic; difficultion; IV fluids indicated 424 platered GI function; tube feeding. FPN or hospitalization indicated; non-emergent operative intervention indicated Definition: A disorder characterized by blockage of the normal flow of the contents of the gallbladder. Gallbladder pain Mild pain Moderate pain; limiting perturn on the discomfort in the gallbladder region. Gallbladder perforation - Life-threatening consequences; Death region. Gallbladder perforation - Life-threatening consequences; Death limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the gallbladder region. Gallbladder perforation - Asterixis; mild encephalopathry; Imiting self care ADL Hepatic failure - Asterixis; mild encephalopathry; Imiting self care ADL intervention indicated by a rupture in the gallbladder wall. Hepatic failure - Asterixis; mild encephalopathry; Imiting self care ADL intervention indicated by the inability of the liver to metabolize chemicals in the body. Laboratory test results reveal abnormal plasma levels of ammonia, bilirubin, lac dehydrogenase, and alkaline phosphalase. Hepatic hemorrhage Mild; intervention not indicated Definition: A disorder characterized by bleeding from the liver. Hepatic necrosis Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent radiologic or operative intervention indicated Definition: A disorder characterized by a necrotic process occurring in the hepatic parenchyma. Hepatic pain intervention indicated Life-threatening consequences; urgent radiologic or operative intervention ind | Definition: A disorder character | rized by an abnormal communication | n between the gallbladder and and | other organ or anatomic site. | | |
| Asymptomatic; clinical or diagnostic observations only; intervention not indicated severally intervention not indicated severally intervention not indicated severally intervention not indicated severally intervention not indicated severally intervention indicated severally intervention indicated severally intervention indicated severally intervention indicated severally intervention indicated severally | Gallbladder necrosis | - | - | - | urgent radiologic or operative | Death |
| diagnostic observations only; intervention not indicated hrs | Definition: A disorder character | rized by a necrotic process occurring | g in the gallbladder. | | | |
| Gallbladder pain Mild pain Moderate pain; limiting instrumental ADL Activities and DL Adsorder characterized by a sensation of marked discomfort in the gallbladder region. Gallbladder perforation Life-threatening consequences; urgent intervention indicated urgent intervention in | | diagnostic observations only;<br>intervention not indicated | function; IV fluids indicated <24 hrs | altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | urgent operative intervention | Death |
| Definition: A disorder characterized by a sensation of marked discomfort in the gallbladder region. Gallbladder perforation Life-threatening consequences; urgent intervention indicated Definition: A disorder characterized by a rupture in the gallbladder wall. Hepatic failure - Asterixis; mild encephalopathy; limiting self care ADL life-threatening consequences; urgent intervention indicated Death limiting self care ADL life-threatening consequences; urgent intervention indicated line threatening consequences. In the body. Laboratory test results reveal abnormal plasma levels of ammonia, billirubin, lace dehydrogenase, and alkaline phosphatase. Hepatic hemorrhage Mild; intervention not indicated line threatening indicated line threatening indicated line threatening consequences; urgent intervention indicated urgent radiologic or operative intervention indicated Definition: A disorder characterized by a necrotic process occurring in the hepatic parenchyma. Hepatic pain Mild pain Moderate pain; limiting limiting limiting limiting liniting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention urgent perative intervention. | | | | | | 1 |
| Definition: A disorder characterized by a rupture in the gallbladder wall. Hepatic failure - Asterixis; mild encephalopathy; limiting self care ADL mechanisms levels of ammonia, bilirubin, lac dehydrogenase, and alkaline phosphatase. Hepatic hemorrhage Mild; intervention not indicated Symptomatic; medical intervention indicated Definition: A disorder characterized by bleeding from the liver. Hepatic necrosis | Gallbladder pain | Mild pain | | | - | - |
| Definition: A disorder characterized by a rupture in the gallbladder wall. Hepatic failure - Asterixis; mild encephalopathy; limiting self care ADL imiting self care ADL imiting self care ADL imiting consequences; urgent intervention indicated intervention: A disorder characterized by the inability of the liver to metabolize chemicals in the body. Laboratory test results reveal abnormal plasma levels of ammonia, bilirubin, lace dehydrogenase, and alkaline phosphatase. Hepatic hemorrhage Mild; intervention not indicated Symptomatic; medical intervention indicated Definition: A disorder characterized by bleeding from the liver. Hepatic necrosis - Life-threatening consequences; urgent radiologic or operative intervention indicated Definition: A disorder characterized by a necrotic process occurring in the hepatic parenchyma. Hepatic pain Mild pain Moderate pain; limiting intervention self-care ADL Severe pain; limiting self care ADL Life-threatening consequences; urgent radiologic or operative intervention indicated - ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention | Definition: A disorder character | rized by a sensation of marked disco | omfort in the gallbladder region. | | | |
| Hepatic failure - Asterixis; mild encephalopathy; limiting self care ADL - Asterixis; mild encephalopathy; limiting self care ADL - Asterixis; mild encephalopathy; limiting self care ADL - Moderate to severe encephalopathy; coma; life-threatening consequences - Definition: A disorder characterized by the inability of the liver to metabolize chemicals in the body. Laboratory test results reveal abnormal plasma levels of ammonia, bilirubin, lac dehydrogenase, and alkaline phosphatase. Hepatic hemorrhage Mild; intervention not indicated Symptomatic; medical intervention indicated Symptomatic; medical intervention indicated Symptomatic; medical intervention indicated Definition: A disorder characterized by bleeding from the liver. Hepatic necrosis Life-threatening consequences; urgent radiologic or operative intervention indicated Definition: A disorder characterized by a necrotic process occurring in the hepatic parenchyma. Hepatic pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention urgent operative intervention | Gallbladder perforation | - | - | - | | Death |
| Definition: A disorder characterized by the inability of the liver to metabolize chemicals in the body. Laboratory test results reveal abnormal plasma levels of ammonia, bilirubin, lac dehydrogenase, and alkaline phosphatase. Hepatic hemorrhage Mild; intervention not indicated Symptomatic; medical intervention indicated intervention indicate | Definition: A disorder character | rized by a rupture in the gallbladder | wall. | | | |
| dehydrogenase, and alkaline phosphatase. Hepatic hemorrhage Mild; intervention not indicated surgent intervention indicated surgent radiologic or operative intervention indicated surgent operative intervention surgent operative interv | Hepatic failure | - | - | limiting self care ADL | encephalopathy; coma; life- | Death |
| Hepatic hemorrhage Mild; intervention not indicated symptomatic; medical intervention indicated wirgent radiologic or operative intervention indicated wirgent radiologic or operative intervention indicated wirgent radiologic or operative intervention indicated wirgent radiologic or operative intervention indicated wirgent radiologic or operative intervention indicated wirgent pain wirgent radiologic or operative intervention indicated wirgent pain | | | etabolize chemicals in the body. L | aboratory test results reveal abnor | mal plasma levels of ammonia, bi | lirubin, lac |
| Hepatic necrosis - Life-threatening consequences; urgent radiologic or operative intervention indicated Definition: A disorder characterized by a necrotic process occurring in the hepatic parenchyma. Hepatic pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention Life-threatening consequences; urgent operative intervention Death - Death | | | | Transfusion indicated | | Death |
| Definition: A disorder characterized by a necrotic process occurring in the hepatic parenchyma. Hepatic pain Mild pain Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention urgent operative intervention | Definition: A disorder character | rized by bleeding from the liver. | | | | |
| Hepatic pain Mild pain Moderate pain; limiting self care instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention Urgent operative intervention | Hepatic necrosis | - | - | - | urgent radiologic or operative | Death |
| instrumental ADL ADL Definition: A disorder characterized by a sensation of marked discomfort in the liver region. Perforation bile duct - Radiologic, endoscopic or elective operative intervention urgent operative intervention | Definition: A disorder character | rized by a necrotic process occurring | g in the hepatic parenchyma. | | | |
| Perforation bile duct - Radiologic, endoscopic or elective operative intervention Life-threatening consequences; urgent operative intervention | Hepatic pain | Mild pain | , , | | - | - |
| elective operative intervention urgent operative intervention | Definition: A disorder character | rized by a sensation of marked disco | omfort in the liver region. | _ | | |
| | Perforation bile duct | - | - | elective operative intervention | urgent operative intervention | Death |

| | | Hepatobiliary diso | rders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Portal hypertension | - | Decreased portal vein flow | Reversal/retrograde portal vein flow; associated with varices and/or ascites | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an increase in blood pressu | re in the portal venous system. | | | |
| Portal vein thrombosis | - | Intervention not indicated | Medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by the formation of a thrombus | (blood clot) in the portal vein. | | | |
| Hepatobiliary disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| | | Immune system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Allergic reaction | Transient flushing or rash, drug fever <38 degrees C (<100.4 degrees F); intervention not indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an adverse local or general | response from exposure to an alle | | | |
| Anaphylaxis | - | - | Symptomatic bronchospasm, with or without urticaria; parenteral intervention indicated; allergy-related edema/angioedema; hypotension | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an acute inflammatory react<br>resents with breathing difficulty, di | • | | | ypersensitivi |
| Autoimmune disorder | | | | | Dooth |
| Autoimmune disorder | Asymptomatic; serologic or<br>other evidence of autoimmune<br>reaction, with normal organ<br>function; intervention not<br>indicated | Evidence of autoimmune reaction involving a non-essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder resulting fr | om loss of function or tissue destru | iction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individe | ual to his ow |
| Cytokine release syndrome | Mild reaction; infusion interruption not indicated; intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for <=24 hrs | following initial improvement;<br>hospitalization indicated for<br>clinical sequelae (e.g., renal<br>impairment, pulmonary<br>infiltrates) | Life-threatening consequences;<br>pressor or ventilatory support<br>indicated | Death |
| Definition: A disorder characteriz | red by nausea, headache, tachyca | rdia, hypotension, rash, and shorti | ness of breath; it is caused by the | release of cytokines from the cells | |
| Serum sickness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate arthralgia; fever, rash, urticaria, antihistamines indicated | Severe arthralgia or arthritis;<br>extensive rash; steroids or IV<br>fluids indicated | Life-threatening consequences; pressor or ventilatory support indicated | Death |
| | red by a delayed-type hypersensiti<br>e foreign antigen. Symptoms inclu | | | | |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the abdominal cavity. | | T | |
| Anorectal infection | Localized; local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | ving the anal area and the rectum. | IV antibiotic antifungal or | Life threatening consequences: | Death |
| Appendicitis | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Deam |
| | rized by acute inflammation to the | | 1 | | ъ " |
| Appendicitis perforated | - | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by acute inflammation to the viceal wall rupture causes the releas | vermiform appendix caused by a pa | athogenic agent with gangrenous o | changes resulting in the rupture of | the |
| Arteritis infective | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving an artery. | | | |
| Biliary tract infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the biliary tract. | 1 | ı | ı |
| Bladder infection | - | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bladder. | | | |
| Bone infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | | T | | |
| Breast infection | - | Local infection with moderate<br>symptoms; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | Severe infection; axillary<br>adenitis; IV antibacterial,<br>antifungal, or antiviral<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | rized by an infectious process invol | 1 | | T | L |
| Bronchial infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process invol | ving the bronchi. | 1 | 1 | 1 |
| Catheter related infection | - | Localized; local intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an infectious process that | arises secondary to catheter use. | | | |
| Cecal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | ed by an infectious process involv | | , and the second | 7 | |
| Cervicitis infection | ed by an incollede process involv | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Cervicius imecuon | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | Death |
| | | antifungal, or antiviral) | radiologic or operative | g | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the uterine cervix. | | | |
| Conjunctivitis infective | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| | | | intervention indicated | 1 | l |
| | ed by an infectious process involv | ring the conjunctiva. Clinical manifo | · · | | I |
| Corneal infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, antifungal, or antiviral) | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | |
| | | and and an animal | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the cornea. | 1 | 1 | • |
| Cranial nerve infection | - '- | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring a cranial nerve. | | | ı |
| Device related infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic or operative | | |
| | | | intervention indicated | 1 | l |
| | ed by an infectious process involv | T | T | I | I |
| Duodenal infection | - | Moderate symptoms; medical | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | intervention indicated (e.g., oral antibiotics) | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | |
| | | 4.142.54.55) | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the duodenum. | ' | • | • |
| Encephalitis infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | severe changes in mental | | |
| | | | status; self-limited seizure | | |
| | | | activity; focal neurologic | | |
| | | 1 | abnormalities | 1 | l |
| | ed by an infectious process involv | ring the brain tissue. | | I | I |
| Encephalomyelitis infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | |
| | | | intervention indicated | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ।<br>ring the brain and spinal cord tissu | 1 | 1 | 1 |
| Endocarditis infective | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | 20001 |
| | | | radiologic or operative | | |
| | | | intervention indicated | | |
| | Ų. | | | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the endocardial layer of the he | eart. | | |
| Definition: A disorder characteriz | ed by an infectious process involv | ring the endocardial layer of the he | Systemic intervention or | Blindness (20/200 or worse) | T- |

| | | Infections and infes | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Enterocolitis infectious | | Passage of >3 unformed stools | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Litteroconus imectious | | per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal | antiviral intervention indicated; radiologic, endoscopic, or | urgent intervention indicated | Deau |
| | | pain | operative intervention indicated;<br>profuse watery diarrhea with<br>signs of hypovolemia; bloody | | |
| | | | diarrhea; fever; severe<br>abdominal pain; hospitalization<br>indicated | | |
| Definition: A disorder characteri | <br>zed by an infectious process involv | ing the small and large intestines | Indicated | | I |
| Esophageal infection | _ | Local intervention indicated | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| Looping Gai milooton | | (e.g., oral antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic or operative | urgent intervention indicated | Dodan |
| | | | intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the esophagus. | T | | |
| Eye infection | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated; | |
| | | antifungal, or antiviral) | radiologic or operative intervention indicated | enucleation | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the eye. | T | Γ | 1 |
| Gallbladder infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | | antiviral intervention indicated; | urgent intervention indicated | |
| | | | radiologic, endoscopic, or operative intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the gallbladder. | | | |
| Gum infection | Local therapy indicated (swish | Moderate symptoms; oral | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | and swallow) | intervention indicated (e.g., | antiviral intervention indicated; | urgent intervention indicated | |
| | | antibiotic, antifungal, antiviral) | radiologic or operative intervention indicated | | |
| Definition: A disorder characteri | zed by an infectious process involv | ing the gums. | T | | |
| Hepatic infection | - | - | IV antibiotic, antifungal, or antiviral intervention indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | radiologic or operative intervention indicated | urgent intervention indicated | |
| Definition: A disorder characteri | l<br>zed by an infectious process involv | I<br>ing the liver | Intervention indicated | l | I |
| Hepatitis viral | Asymptomatic, treatment not | - | Symptomatic liver dysfunction; | Decompensated liver function | Death |
| | indicated | | fibrosis by biopsy; compensated cirrhosis; reactivation of chronic hepatitis | (e.g., ascites, coagulopathy, encephalopathy, coma) | |
| Definition: A disorder characteri | ।<br>zed by a viral pathologic process ir | l<br>volving the liver parenchyma | Inopatito | Į. | 1 |
| Infective myositis | - | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| • | | indicated (e.g., topical antibiotic, | antiviral intervention indicated; | urgent intervention indicated | |
| | | antifungal, or antiviral) | radiologic or operative | | |
| Definition: A disorder characteri | <br>zed by an infectious process involv | ing the skeletal muscles | intervention indicated | I | I |
| Joint infection | - | Localized; local intervention | Arthroscopic intervention | Life-threatening consequences; | Death |
| | | indicated; oral intervention | indicated (e.g., drainage) or | urgent intervention indicated | |
| | | indicated (e.g., antibiotic, | arthrotomy (e.g., open surgical | | |
| | | antifungal, antiviral); needle | drainage) | | |
| | | aspiration indicated (single or multiple) | | | |
| Definition: A disorder characteri | ।<br>zed by an infectious process involv | | ı | I | I |
| Kidney infection | - | - | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| • | | | antiviral intervention indicated; | urgent intervention indicated | 1 |
| | | | radiologic, endoscopic, or | | |
| | | | operative intervention indicated | | 1 |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by an inflammatory process i | nvolving the larynx. | | | |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder charac | cterized by an infectious process invo | lving the lips. | | | |
| Lung infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by an infectious process invo | lving the lungs. | T | T | I |
| Lymph gland infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | cterized by an infectious process invo | lving the lymph nodes. | I | 1 | |
| Mediastinal infection | | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by an infectious process invo | lving the mediastinum. | 1 | 1 | |
| Meningitis | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by acute inflammation of the | meninges of the brain and/or spinal | cord. | 1 | · · |
| Mucosal infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by an infectious process invo | lving a mucosal surface. | | | |
| Nail infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder charac | cterized by an infectious process invo | lving the nail. | T | T | |
| Otitis externa | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | cterized by an infectious process invo<br>ymptoms include fullness, itching, swe | • | • | ive water exposure (swimmer's ea | r infectior |
| Otitis media | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by an infectious process invo | lving the middle ear. | | · | |
| Ovarian infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative | Life-threatening consequences; urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involv | ing the pancreas. | | | |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | erized by an eruption consisting of pa | | | | o, and upper |
| | this rash does not present with whiteh | | İ | esions. | |
| Paronychia | Nail fold edema or erythema;<br>disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical intervention or IV antibiotics indicated; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by an infectious process involvi | ing the soft tissues around the nai | ļ. | | |
| Pelvic infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by an infectious process involving | ing the pelvic cavity. | <u> </u> | 1 | |
| Penile infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involvi | ing the penis. | | | |
| Periorbital infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by an infectious process involvi | | D/ | if_ | D41- |
| Peripheral nerve infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by an infectious process involvi | ing the peripheral nerves. | | | |
| Peritoneal infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process involvi | ing the peritoneum. | 1 | 1 | |
| Pharyngitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by inflammation of the throat. | ·<br> | | | |
| Phlebitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz of the infected vein. | ed by an infectious process involvi | ing the vein. Clinical manifestation | s include erythema, marked disco | mfort, swelling, and induration alo | ng the course |
| Pleural infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the pleura. | | | |
| Prostate infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the prostate gland. | I | I | |
| Rash pustular | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a circumscribed and elevate | d skin lesion filled with pus. | T | T | 1 |
| Rhinitis infective | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | - | - | - |
| | ed by an infectious process involvi | | In | | |
| Salivary gland infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the salivary gland. | | | |
| Scrotal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the scrotum. | T | T | 1 |
| Sepsis | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by the presence of pathogenic | microorganisms in the blood strea | m that cause a rapidly progressin | g systemic reaction that may lead | to shock. |
| Sinusitis | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the mucous membranes of the | paranasal sinuses. | T | |
| Skin infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the skin. | T | T | T |
| Small intestine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an infectious process involvi | ing the small intestine. | T | T | |
| Soft tissue infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by an infectious process involvi | ing soft tissues. | | I | I |
| Splenic infection | - | - | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | ized by an infectious process involv | | v | 7 | |
| Stoma site infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing a stoma (surgically created op | ening on the surface of the body). | 1 | |
| Tooth infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing a tooth. | T | 1 | 1 |
| Tracheitis | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ized by an infectious process involv | | | | I |
| Upper respiratory infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the upper respiratory tract (nos | se, paranasal sinuses, pharynx, la | rynx, or trachea). | ı |
| Urethral infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the urethra. | | | |
| Urinary tract infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the urinary tract, most commo | nly the bladder and the urethra. | • | · |
| Uterine infection | - | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the endometrium. It may exten | ,<br>d to the myometrium and parame | trial tissues. | • |
| Vaginal infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the vagina. | 1 | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the vulva. | | | |
| Wound infection | - | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the wound. | | 1 | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Injury, poisoning and procedural complications Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention | Limiting instrumental ADL; | Limiting self care ADL; elective | - <del>-</del> | _ |
| | indicated | operative intervention indicated | surgery indicated | | |
| Definition: A finding of damage in<br>Affected leg and foot. | to the ankle joint characterized by a | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | y moving th |
| Aortic injury | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | | | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage | to the aorta. | 1 | | l | |
| Arterial injury | Asymptomatic diagnostic | Symptomatic (e.g., | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| , , | finding; intervention not indicated | claudication); repair or revision not indicated | care ADL; disabling; repair or revision indicated | evidence of end organ damage;<br>urgent operative intervention<br>indicated | |
| Definition: A finding of damage | to an artery. | | | • | |
| Biliary anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | | |
| Deficitions A finalism of locks | not indicated | | intervention indicated | indicated | l |
| | of bile due to breakdown of a biliary | | | | D4h |
| Bladder anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | of urine due to breakdown of a blad | dder anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | |
| Bruising | Localized or in a dependent area | Generalized | - | - | - |
| Definition: A finding of injury of t | he soft tissues or bone characteriz | ed by leakage of blood into surrou | nding tissues. | | 1 |
| Burn | Minimal symptoms; intervention not indicated | Medical intervention; minimal debridement indicated | Moderate to major debridement or reconstruction indicated | Life-threatening consequences | Death |
| • . | integrity to the anatomic site of an depends on the length and intensi | | * * | nicals, direct heat, electricity, flame | es and |
| Dermatitis radiation | Faint erythema or dry | Moderate to brisk erythema; | Moist desquamation in areas | Life-threatening consequences; | Death |
| Joinnaulo radiation | desquamation | patchy moist desquamation, | other than skin folds and | skin necrosis or ulceration of full | Boati |
| | | mostly confined to skin folds | creases; bleeding induced by | thickness dermis; spontaneous | |
| | | and creases; moderate edema | minor trauma or abrasion | bleeding from involved site; skin graft indicated | |
| Definition: A finding of cutaneou | <br> s inflammatory reaction occurring a | <br>as a result of exposure to biologica | I<br>Illy effective levels of ionizing radia | 19 | I |
| Esophageal anastomotic leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| _sopriageal anastomotic leak | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | ।<br>due to breakdown of an esophagea | l anastomosis (surgical connection | ।<br>n of two separate anatomic structu | res). | |
| Fall | Minor with no resultant injuries; intervention not indicated | Symptomatic; noninvasive intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding of sudden n | novement downward, usually result | ting in injury. | , | | |
| Fallopian tube anastomotic leak | Asymptomatic; clinical or | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | |
| Definition: A finding of leakage of | due to breakdown of a fallopian tub | e anastomosis (surgical connectio | n of two separate anatomic structu | ıres). | |
| Fallopian tube perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture o | f the fallopian tube wall. | 1 | | | |
| Fracture | Asymptomatic; clinical or | Symptomatic but non-displaced; | Severe symptoms; displaced or | Life-threatening consequences; | Death |
| | diagnostic observations only; intervention not indicated | immobilization indicated | open wound with bone exposure; disabling; operative | urgent intervention indicated | |

| Injury, poisoning and procedural complications Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic observations only; intervention | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative | Life-threatening consequences; urgent operative intervention | Death |
| | not indicated | Intervention indicated | intervention indicated | indicated | |
| Deficialization of localization of | 1 | <br>+ | • | Indicated | l |
| | | tomosis (surgical connection of tw | | T | I |
| Gastrointestinal anastomotic | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| leak | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | I | intervention indicated | indicated | |
| Definition: A finding of leakage d | ue to breakdown of a gastrointesti | nal anastomosis (surgical connect | tion of two separate anatomic struc | ctures). | |
| Gastrointestinal stoma necrosis | - | Superficial necrosis; | Severe symptoms; | Life-threatening consequences; | Death |
| | | intervention not indicated | hospitalization or elective | urgent intervention indicated | |
| | | | operative intervention indicated | | |
| Definition: A finding of a necrotic | process occurring in the gastroint | estinal tract stoma. | | | |
| Hip fracture | - | Hairline fracture; mild pain; | Severe pain; hospitalization or | Life-threatening consequences; | - |
| | | limiting instrumental ADL; non- | intervention indicated for pain | symptoms associated with | |
| | | surgical intervention indicated | control (e.g., traction); operative | neurovascular compromise | |
| | | | intervention indicated | | |
| Definition: A finding of traumatic | injury to the hip in which the contii | nuity of either the femoral head, fe | moral neck, intertrochanteric or su | btrochanteric regions is broken. | |
| Injury to carotid artery | - | - | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| to our old artory | | | care ADL (e.g., transient | urgent intervention indicated | Dogui |
| | | | cerebral ischemia); repair or | January Straight Middled | |
| | | | revision indicated | | |
| Definition: A finding of damage to | the carotid artery | ı | 1 | ı | 1 |
| Injury to inferior vena cava | | | | Life threatening consequences: | Death |
| injury to intenor vena cava | - | - | - | Life-threatening consequences; urgent intervention indicated | Dealii |
| | | 1 | I | urgent intervention indicated | l |
| Definition: A finding of damage to | the interior vena cava. | 1 | | Τ | 1 |
| Injury to jugular vein | - | - | Symptomatic limiting self care | Life-threatening consequences; | Death |
| | | | ADL; disabling; repair or | urgent intervention indicated | |
| | I | I | revision indicated | I | |
| Definition: A finding of damage to | the jugular vein. | 1 | 1 | T | |
| Injury to superior vena cava | Asymptomatic diagnostic | Symptomatic; repair or revision | Severe symptoms; limiting self | Life-threatening consequences; | Death |
| | finding; intervention not | not indicated | care ADL; disabling; repair or | evidence of end organ damage; | |
| | indicated | | revision indicated | urgent operative intervention | |
| | | | 1 | indicated | |
| Definition: A finding of damage to | the superior vena cava. | | | | |
| Intestinal stoma leak | Asymptomatic diagnostic | Symptomatic; medical | Severe symptoms; radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention | intervention indicated | endoscopic or elective operative | urgent operative intervention | |
| | not indicated | | intervention indicated | indicated | |
| Definition: A finding of leakage of | contents from an intestinal stoma | a (surgically created opening on th | e surface of the body). | | |
| Intestinal stoma obstruction | - | Self-limited; intervention not | Severe symptoms; IV fluids, | Life-threatening consequences; | Death |
| | | indicated | tube feeding, or TPN indicated | urgent operative intervention | |
| | | | >=24 hrs; elective operative | indicated | |
| | | | intervention indicated | | |
| Definition: A finding of blockage | of the normal flow of the contents | of the intestinal stoma. | • | • | • |
| Intestinal stoma site bleeding | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| mostinai stoma site biecuilly | clinical exam; intervention not | intervention indicated | indicated; radiologic or | urgent intervention indicated | Doani |
| | indicated | | endoscopic intervention | a.g.s.ik intorvontion indicated | |
| | | | indicated | | |
| Definition: A finding of blood leak | age from the intestinal stoma | 1 | 1 | I | 1 |
| | | D 01 0 01 1 | 0 11 " | Lee al | D .: |
| Intraoperative arterial injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| | organ/structure indicated | organ/structure indicated | reconstruction of injured | urgent intervention indicated | |
| | | | organ/structure indicated; | | |
| <b>.</b> | l | | disabling | I | I |
| Definition: A finding of damage to | o an artery during a surgical proce | dure. | | <u> </u> | |
| Intraoperative breast injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| | organ/structure indicated | organ/structure indicated | reconstruction of injured | urgent intervention indicated | |
| | į. | ĺ | lorgon/structure indicated: | İ | 1 |
| | | | organ/structure indicated; disabling | | |

| | | , poisoning and proced | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | o the breast parenchyma during a | | • | <del>-</del> | |
| Intraoperative cardiac injury | - | - | Primary repair of injured organ/structure indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the heart during a surgical proce | edure. | | | |
| Intraoperative ear injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection of injured organ/structure indicated; disabling (e.g., impaired hearing; impaired balance) | Life-threatening consequences; urgent intervention indicated | Death |
| | o the ear during a surgical proced | | | | I |
| Intraoperative endocrine injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the endocrine gland during a sui | rgical procedure. | | | |
| Intraoperative gastrointestinal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the gastrointestinal system durin | g a surgical procedure. | | | |
| Intraoperative head and neck<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the head and neck during a surg | ical procedure. | | | |
| Intraoperative hemorrhage | - | - | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical proc | edure. | ı | ! | • |
| Intraoperative hepatobiliary injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the hepatic parenchyma and/or | biliary tract during a surgical pro | cedure. | | |
| Intraoperative musculoskeletal<br>injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the musculoskeletal system duri | ng a surgical procedure. | | | |
| Intraoperative neurological injury | Primary repair of injured organ/structure indicated of the nervous system during a sur | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | | Ĭ | 0 11 " | | Б. " |
| Intraoperative ocular injury | Primary repair of injured organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the eye during a surgical proced | ure. | | | |
| Intraoperative renal injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | o the kidney during a surgical prod | cedure. | ·<br> | · | |
| Intraoperative reproductive tract injury | | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| Injury, poisoning and procedural complications Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | the reproductive organs during a | | | · | |
| Intraoperative respiratory injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the respiratory system during a s | surgical procedure. | | | |
| Intraoperative skin injury | Primary repair of injured organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the skin during a surgical proced | ure. | | | |
| Intraoperative splenic injury | the prices during a surgical president | Primary repair of injured organ/structure indicated | Resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| | the spleen during a surgical proc | | Complete resection or | Life threatening concernance | Dooth |
| Intraoperative urinary injury Definition: A finding of damage to | Primary repair of injured organ/structure indicated the urinary system during a surg | Partial resection of injured organ/structure indicated ical procedure. | Complete resection or reconstruction of injured organ/structure indicated; disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Intraoperative venous injury | Primary repair of injured | Partial resection of injured | Complete resection or | Life-threatening consequences; | Death |
| muaoperauve venous injury | organ/structure indicated | organ/structure indicated | reconstruction of injured organ/structure indicated; disabling | urgent intervention indicated | Deali |
| Definition: A finding of damage to | a vein during a surgical procedu | re. | · | | |
| Kidney anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | urine due to breakdown of a kidn | ey anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage du | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| <u> </u> | · · | nastomosis (surgical connection o | T ' | Í | 1 |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | indicated | Death |
| | | anastomosis (surgical connection | | ľ | |
| Postoperative hemorrhage | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; radiologic, endoscopic, or operative intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics) pRBCs beyond protocol specification; urgent radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ccurring after a surgical procedur | | Figure 4 and 5 70 f | I the share to the | D |
| Postoperative thoracic procedure complication | - | Extubated within 24 - 72 hrs postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A finding of a previous | ly undocumented problem that oc | curs after a thoracic procedure. | 1 | I | |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental | Severe symptoms; elective operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent operative intervention indicated | Death |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of protrusion | of the intestinal stoma (surgically | created opening on the surface of | the body) above the abdominal s | urface. | |
| Prolapse of urostomy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective operative intervention or major stomal revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of displacem | ent of the urostomy. | | | | |
| Radiation recall reaction<br>(dermatologic) | Faint erythema or dry desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| | inflammatory reaction caused by | | - | owing radiotherapy. The inflamma | tory react |
| · | liated skin and the symptoms disa | i · | I . | | |
| Rectal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a rectal anasto | omosis (surgical connection of two | separate anatomic structures). | | Г |
| Seroma | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; simple aspiration indicated | Symptomatic, elective radiologic or operative intervention indicated | - | - |
| Definition: A finding of tumor-like | collection of serum in the tissues. | T | T | Г | |
| Small intestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an anastomos | is (surgical connection of two sepa | arate anatomic structures) in the si | mall bowel. | |
| Spermatic cord anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a spermatic co | ord anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Spinal fracture | Mild back pain; nonprescription analgesics indicated | Moderate back pain;<br>prescription analgesics<br>indicated; limiting instrumental<br>ADL | Severe back pain;<br>hospitalization or intervention<br>indicated for pain control (e.g.,<br>vertebroplasty); limiting self care<br>ADL; disability | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise | Death |
| Definition: A finding of traumatic | injury to the spine in which the cor | ntinuity of a vertebral bone is broke | en. | ! | • |
| Stenosis of gastrointestinal stoma | of the gastrointestinal stome (sur | Symptomatic; IV fluids indicated <24 hrs; manual dilation at bedside | tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | of the gastrointestinal stoma (surg | | | | |
| Stomal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by a circumscribed, inflammato | ory and necrotic erosive lesion on t | the jejunal mucosal surface close t | to the anastomosis site following a | |
| Tracheal hemorrhage | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| v | clinical or diagnostic exam;<br>intervention not indicated | intervention indicated | indicated; radiologic or<br>endoscopic intervention<br>indicated | urgent intervention indicated | |
| Definition: A finding of bleeding f | | | T. | | |
| Tracheal obstruction | Partial asymptomatic<br>obstruction on examination<br>(e.g., visual, radiologic or<br>endoscopic) | Symptomatic (e.g., noisy airway breathing), no respiratory distress; medical intervention indicated (e.g., steroids); limiting | Stridor; radiologic or endoscopic intervention indicated (e.g., stent, laser); limiting self care ADL | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |

| Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Tracheostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of blood lea | kage from the tracheostomy site. | + | | | |
| Ureteric anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic, endoscopic or elective operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | lue to breakdown of a ureteral ana | T T | | T . | |
| Jrethral anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a urethral ana | stomosis (surgical connection of tw | vo separate anatomic structures). | | |
| Urostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | of contents from a urostomy. | 1 | 1 | T | |
| Urostomy obstruction | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; dilation or<br>endoscopic repair or stent<br>placement indicated | Altered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | | | | |
| Urostomy site bleeding | Minimal bleeding identified on clinical exam; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of bleeding | from the urostomy site. | ' | ' | ' | • |
| Urostomy stenosis | - | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g.,<br>hydronephrosis, or renal<br>dysfunction); elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of narrowing | g of the opening of a urostomy. | | | | |
| Uterine anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a uterine anas | tomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a rupture in the uterine wall. | | 0 | | D41- |
| /aginal anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage o | lue to breakdown of a vaginal anas | stomosis (surgical connection of tw | o separate anatomic structures). | | 1 |
| /as deferens anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vas deferens | s anastomosis (surgical connection | n of two separate anatomic structu | res). | |
| Vascular access complication | - | Device dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including pulmonary embolism or life-threatening thrombus | Death |

| | Injury | , poisoning and procedu | ral complications | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Venous injury | Asymptomatic diagnostic finding; intervention not indicated | Symptomatic (e.g., claudication); repair or revision not indicated | Severe symptoms; limiting self<br>care ADL; repair or revision<br>indicated; disabling | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | a vein. | | | | |
| Wound complication | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound; local care indicated | Hernia without evidence of<br>strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by<br>operative intervention indicated | Hernia with evidence of<br>strangulation; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| · · · · · · | Incisional separation of <=25% | 1 | Fascial disruption or dehiscence | Life threatening concessions | Dooth |
| Wound dehiscence | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of wound with local care; asymptomatic hernia or symptomatic hernia without evidence of strangulation | Hascial disruption or deniscence without evisceration; primary wound closure or revision by operative intervention indicated | Life-threatening consequences; symptomatic hernia with evidence of strangulation; fascial disruption with evisceration; major reconstruction flap, grafting, resection, or amputation indicated | Death |
| Definition: A finding of separation | of the approximated margins of a | surgical wound. | T | Г | 1 |
| Wrist fracture | Mild; non-surgical intervention indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | - | - |
| Definition: A finding of traumatic | injury to the wrist joint in which the | continuity of a wrist bone is broke | en. | | |
| Injury, poisoning and procedural complications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Investigations | <b>S</b> | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | y test result in which the partial th | | | possible indicator of coagulopat | hy, a prolonge |
| , , | may occur in a variety of disease | | | | |
| Alanine aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | | 1 , | 1 | 1 |
| Alkaline phosphatase increased | 1 | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | · | · | | |
| Aspartate aminotransferase increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen. | _ |
| Blood antidiuretic hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of antidiuretic horm | one in the blood specimen. | | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is as | ssociated with jaundice. | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotropl | nin in a blood specimen. | | |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; | Symptomatic; medical intervention indicated; limiting instrumental ADI | Severe symptoms; limiting self care ADL | - | - |
| Definition A finding board on lab | intervention not indicated | instrumental ADL | | | I |
| | oratory test results that indicate a | 1 | ormone in a blood specimen. | | 1 |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | ,<br>bnormal levels of prolactin hormor | ne in a blood specimen. | ' | • |
| Carbon monoxide diffusing capacity decreased | 3 - 5 units below LLN; for follow-<br>up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | 6 - 8 units below LLN; for follow-<br>up, an asymptomatic decrease<br>of >5 - 8 units (ml/min/mm Hg)<br>below the baseline value | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., >Grade 2 hypoxia or >Grade 2 or higher dyspnea) | - | - |
| Definition: A finding based on lun | g function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | ' | • |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| · | t which indicates increased levels | of cardiac troponin I in a biologica | 1 | | 1 |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test resul | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | | ·<br> |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | |
| Cholesterol high | >ULN - 300 mg/dL; >ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL; >10.34 -<br>12.92 mmol/L | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | oratory test results that indicate h | gher than normal levels of cholest | terol in a blood specimen. | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in levels of creatine pho | osphokinase in a blood specimen. | | |

| Investigations | | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5 x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate in | ncreased levels of creatinine in a b | iological specimen. | | |
| Ejection fraction decreased | - | Resting ejection fraction (EF) 50 - 40%; 10 - 19% drop from baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline | Resting ejection fraction (EF) <20% | - |
| Definition: The percentage comp contraction. | uted when the amount of blood ej | ected during a ventricular contract | ion of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected interval prolonged | | QTc 481 - 500 ms | QTc >= 501 ms on at least two separate ECGs | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| Definition: A finding of a cardiac | dysrhythmia characterized by an a<br>r | abnormally long corrected QT inter | val.<br>T | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25%<br>decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <pre>&lt;0.5 - 0.25 x LLN or 50 - &lt;75% decrease from baseline</pre> | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of fibrinogen i | in a blood specimen. | | |
| Forced expiratory volume<br>decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| Definition: A finding based on tes | t results that indicate a relative de | ecrease in the fraction of the forced | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | | - | zyme gamma-glutamyltransferase | | ıma- |
| | | | tide to another peptide, amino acid<br>T | s or water. | |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of growth hormone | in a biological specimen. | | |
| Haptoglobin decreased | <lln< td=""><td>-</td><td>-</td><td>-</td><td>-</td></lln<> | - | - | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of haptoglobin | n in a blood specimen. | | |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN | Increase in >2 - 4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN | - | - |
| Definition: A finding based on lab | oratory test results that indicate in | ncreased levels of hemoglobin in a | biological specimen. | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>anticoagulation | >2.5 x ULN; >2.5 times above baseline if on anticoagulation | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the ratio of the patier | nt's prothrombin time to a control s | ample in the blood. | |
| Lipase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of lipase in | a biological specimen. | | |
| Lymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of lymphocyt | es in a blood specimen. | | |
| Lymphocyte count increased | - | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormal increase in the numbe | r of lymphocytes in the blood, effu | sions or bone marrow. | |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of neutrophils | s in a blood specimen. | | |
| Pancreatic enzymes decreased | <lln and="" asymptomatic<="" td=""><td>Increase in stool frequency, bulk, or odor; steatorrhea</td><td>Sequelae of absorption deficiency</td><td>-</td><td>-</td></lln> | Increase in stool frequency, bulk, or odor; steatorrhea | Sequelae of absorption deficiency | - | - |
| | • | • | • | • | |

| | | Investigations | • | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<br="" 75,000="" <lln="" mm3;="">75.0 x 10e9 /L</lln> | <75,000 - 50,000/mm3; <75.0 - 50.0 x 10e9 /L | <50,000 - 25,000/mm3; <50.0 -<br>25.0 x 10e9 /L | <25,000/mm3; <25.0 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the levels of amylase | e in a serum specimen. | • | • |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | _ |
| Definition: A finding based on tes | t results that indicate urine produc | tion is less relative to previous ou | tput. | • | ` |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value;<br>limiting instrumental ADL | <50% of predicted value;<br>limiting self care ADL | - | - |
| Definition: A finding based on pu value. | Imonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | uum inhalation) when compared to | the predicted |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characterize | d by an increase in overall body w | eight; for pediatrics, greater than t | he baseline growth curve. | | |
| Weight loss | 5 to <10% from baseline;<br>intervention not indicated | 10 - <20% from baseline;<br>nutritional support indicated | >=20% from baseline; tube<br>feeding or TPN indicated | - | - |
| Definition: A finding characterize | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <3000 - 2000/mm3; <3.0 - 2.0 x<br>10e9 /L | <2000 - 1000/mm3; <2.0 - 1.0 x<br>10e9 /L | <1000/mm3; <1.0 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in number of white blo | od cells in a blood specimen. | | |
| Investigations - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| cidosis | pH <normal, but="">=7.3</normal,> | - | pH <7.3 | Life-threatening consequences | Death |
| efinition: A disorder characteriz | zed by abnormally high acidity (high | h hydrogen-ion concentration) of t | he blood and other body tissues. | | |
| Alcohol intolerance | - | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an increase in sensitivity to | the adverse effects of alcohol, wh | ich can include nasal congestion, | skin flushes, heart dysrhythmias, i | nausea, |
| romiting, indigestion and heada<br>Alkalosis | | | pH >7.5 | Life threatening consequences | Dooth |
| | pH >normal, but <=7.5 | <del>-</del><br> | 1. | Life-threatening consequences | Death |
| | zed by abnormally high alkalinity (lo | | | | I <sub>D</sub> ,, |
| Anorexia | Loss of appetite without alteration in eating habits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a loss of appetite. | | | | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | zed by excessive loss of water from | the body. It is usually caused by | severe diarrhea, vomiting or diaph | oresis. | |
| Glucose intolerance | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences; urgent intervention indicated | Death |
| efinition: A disorder characteriz | zed by an inability to properly metal | bolize glucose. | | | |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; lonized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteriz | zed by laboratory test results that ir | ,<br>ndicate an elevation in the concen | ration of calcium (corrected for all | oumin) in blood. | • |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8.9 mmol/L | Fasting glucose value >160 -<br>250 mg/dL; Fasting glucose<br>value >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder characteriz<br>ntolerance. | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of blood sugar. It is usually | an indication of diabetes mellitus | or glucose |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize the use of diuretic drugs. | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of potassium in the blood; a | associated with kidney failure or so | ometimes w |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23<br>mmol/L | - | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that in | ndicate an elevation in the concen | tration of magnesium in the blood | T | |
| lypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characterize | zed by laboratory test results that in | | | T | T |
| lypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | >300 mg/dL - 500 mg/dL; >3.42<br>mmol/L - 5.7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | >1000 mg/dL; >11.4 mmol/L;<br>life-threatening consequences | Death |
| efinition: A disorder characteriz | zed by laboratory test results that in | ndicate an elevation in the concen | | | 1 |
| lyperuricemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | - | >ULN - 10 mg/dL (0.59 mmol/L) with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| efinition: A disorder characteriz | zed by laboratory test results that ir | ndicate an elevation in the concen | tration of uric acid. | 1 | 1 |
| ypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by laboratory test results that ir | ndicate a low concentration of albu | ımin in the blood. | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -<br="">1.0 mmol/L</lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of <7.0 - 6.0 mg/dL; <1.75 - 1.5 mmol/L; lonized calcium <0.9 - 0.8 mmol/L; hospitalization indicated | Corrected serum calcium of <6.0 mg/dL; <1.5 mmol/L; lonized calcium <0.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate a low concentration of calc | ium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0="" 55="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;55 - 40 mg/dL; &lt;3.0 - 2.2<br/>mmol/L</td><td>&lt;40 - 30 mg/dL; &lt;2.2 - 1.7<br/>mmol/L</td><td>&lt;30 mg/dL; &lt;1.7 mmol/L; life-<br/>threatening consequences;<br/>seizures</td><td>Death</td></lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 mg/dL; <1.7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of gluc | cose in the blood. | | |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <lln -="" 3.0="" l;<br="" mmol="">symptomatic; intervention<br/>indicated</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate a low concentration of pota | assium in the blood. | | |
| Hypomagnesemia | <lln -="" 0.5="" 1.2="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;1.2 - 0.9 mg/dL; &lt;0.5 - 0.4 mmol/L</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 - 0.3 mmol/L</td><td>&lt;0.7 mg/dL; &lt;0.3 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <1.2 - 0.9 mg/dL; <0.5 - 0.4 mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3 mmol/L | <0.7 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of mag | gnesium in the blood. | | |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td>-</td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | - | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that in | ndicate a low concentration of sod | ium in the blood. | | |
| Hypophosphatemia | <lln -="" 0.8="" 2.5="" <lln="" dl;="" l<="" mg="" mmol="" td=""><td>&lt;2.5 - 2.0 mg/dL; &lt;0.8 - 0.6 mmol/L</td><td>&lt;2.0 - 1.0 mg/dL; &lt;0.6 - 0.3<br/>mmol/L</td><td>&lt;1.0 mg/dL; &lt;0.3 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6 mmol/L | <2.0 - 1.0 mg/dL; <0.6 - 0.3<br>mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-threatening consequences | Death |
| Definition: A disorder characteri | zed by laboratory test results that ir | ndicate a low concentration of pho | sphates in the blood. | | |
| Iron overload | - | Moderate symptoms; intervention not indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by accumulation of iron in the t | issues. | | _ | |
| Obesity | - | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | - |
| Definition: A disorder characteri | zed by having a high amount of boo | dy fat. | | | |
| Tumor lysis syndrome | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by metabolic abnormalities that | t result from a spontaneous or the | rapy-related cytolysis of tumor cell | s. | |
| Metabolism and nutrition<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal soft tissue necrosis | - | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the abdomir | nal wall. | | |
| Arthralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | mfort in a joint. | T | 1 | Г |
| Arthritis | Mild pain with inflammation, erythema, or joint swelling | Moderate pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by inflammation involving a joir | it. | 1 | 1 | 1 |
| Avascular necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by necrotic changes in the bond<br>and the destruction of the bone struc | | d supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the back region. | | _ | |
| Bone pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the bones. | T | 1 | Г |
| Buttock pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the buttocks. | | | |
| Chest wall pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n in the chest wall region. | T | T | |
| Exostosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated | - | - |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth o | of bone. | • | | |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the | deep connective tissues. | 1 | 1 | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort sensation | n on the lateral side of the body in | the region below the ribs and abo | ove the hip. | 1 |
| Generalized muscle weakness | Symptomatic; weakness<br>perceived by patient but not<br>evident on physical exam | Symptomatic; weakness evident on physical exam; weakness limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | - |
| | ed by a reduction in the strength o | · . | | | |
| Growth suppression | Reduction in growth velocity by 10 - 29% ideally measured over the period of a year ed by of stature that is smaller that | Reduction in growth velocity by 30 - 49% ideally measured over the period of a year or 0 - 49% reduction in growth from the baseline growth curve | Reduction in growth velocity of >=50% ideally measured over the period of a year | - | - |

| Musculoskeletal and connective tissue disorders Grade | | | | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Head soft tissue necrosis | | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a necrotic process occurring | in the soft tissues of the head. | • | • | |
| Joint effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self care ADL; elective operative intervention indicated; disabling | - | - |
| Definition: A disorder characteriz | ed by excessive fluid in a joint, usu | ually as a result of joint inflammation | on. | | |
| Joint range of motion decreased | <=25% loss of ROM (range of<br>motion); decreased ROM<br>limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50% decrease in ROM; limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a decrease in joint flexibility | of any joint. | | | |
| Joint range of motion decreased cervical spine | Mild restriction of rotation or flexion between 60 - 70 degrees | Rotation <60 degrees to right or left; <60 degrees of flexion | Ankylosed/fused over multiple segments with no C-spine rotation | - | - |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | cervical spine joint. | T | T | |
| Joint range of motion decreased lumbar spine | Stiffness; difficulty bending to the floor to pick up a very light object but able to do athletic activity | Pain with range of motion (ROM) in lumbar spine; requires a reaching aid to pick up a very light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>ankylosis or fused over multiple<br>segments with no L-spine<br>flexion (e.g., unable to reach to<br>floor to pick up a very light<br>object) | - | - |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | lumbar spine joint. | | | |
| Kyphosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ·<br>ed by an abnormal increase in the | curvature of the thoracic portion o | of the spine. | • | • |
| Lordosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the lumbar portion of | the spine. | | |
| Muscle weakness left-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the left side of th | e body. | <b>-</b> | |
| Muscle weakness lower limb | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the lower limb muscles. | | <del> </del> | |
| Muscle weakness right-sided | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the right side of t | he body. | T | |
| Muscle weakness trunk | Symptomatic; perceived by patient but not evident on physical exam | Symptomatic; evident on physical exam; limiting instrumental ADL | Limiting self care ADL; disabling | - | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the trunk muscles. | | <b>-</b> | |
| Muscle weakness upper limb | Symptomatic; perceived by | Symptomatic; evident on | Limiting self care ADL; disabling | | - |

| Musculoskeletal and connective tissue disorders | | | | | |
|---|---|---|---|---|---|
| | Grade 1 2 3 4 5 | | | | |
| Adverse Event | 1 | 2 | | 4 | 5 |
| Musculoskeletal deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g.,<br>shoe insert) or covered by<br>clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; disabling | - | - |
| Definition: A disorder characteri | zed by of a malformation of the mu | sculoskeletal system. | | | |
| Myalgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | | |
| Myositis | Mild pain | Moderate pain associated with weakness; pain limiting instrumental ADL | Pain associated with severe weakness; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by inflammation involving the s | keletal muscles. | | | |
| Neck pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the neck area. | T | | T |
| Neck soft tissue necrosis | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | g in the soft tissues of the neck. | | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of<br>osteoporosis or Bone Mineral<br>Density (BMD) t-score -1 to -2.5<br>(osteopenia); no loss of height<br>or intervention indicated | BMD t-score <-2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm;<br>hospitalization indicated; limiting<br>self care ADL | - | - |
| Definition: A disorder characteri composition), resulting in increa | zed by reduced bone mass, with a used fracture incidence. | decrease in cortical thickness and | in the number and size of the trab | peculae of cancellous bone (but no | ormal chemi |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the upper or lower extremities | ·<br>i. | | |
| Pelvic soft tissue necrosis | - zed by a necrotic process occurring | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Scoliosis | <20 degrees; clinically | | >45 dogrado: acopular | | |
| SCOIIOSIS | undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | | - |
| Definition: A disorder characteri | zed by a malformed, lateral curvatu | re of the spine. | 1 | <u> </u> | |
| Soft tissue necrosis lower limb | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | g in the soft tissues of the lower ex | tremity. | 1 | |
| Soft tissue necrosis upper limb | - | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other invasive intervention indicated (e.g., tissue reconstruction, flap or grafting) | Life-threatening consequences; urgent intervention indicated | Death |

| | Musculoskeletal and connective tissue disorders | | | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superficial soft tissue fibrosis | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| Definition: A disorder characterize | ed by fibrotic degeneration of the s | superficial soft tissues. | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, soft foods or purees | Decreased ROM with inability to adequately aliment or hydrate orally | - | - |
| Definition: A disorder characterize | ed by lack of ability to open the mo | outh fully due to a decrease in the | range of motion of the muscles of | mastication. | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 - 5 cm; shoe lift indicated; limiting instrumental ADL | | - | - |
| Definition: A disorder characterize | ed by of a discrepancy between th | e lengths of the lower or upper ex | tremities. | | |
| Musculoskeletal and connective tissue disorder - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Neoplasms benig | n, malignant and unspec | cified (incl cysts and poly | yps) | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Leukemia secondary to oncology chemotherapy | - | - | - | Present | Death |
| Definition: A disorder characterize | ed by leukemia arising as a result | of the mutagenic effect of chemot | herapy agents. | | |
| Myelodysplastic syndrome | - | - | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by insufficiently healthy hemata | poietic cell production by the bone | e marrow. | | |
| Treatment related secondary malignancy | - | - | Non life-threatening secondary malignancy | Acute life-threatening secondary malignancy; blast crisis in leukemia | Death |
| Definition: A disorder characterize | ed by development of a malignand | by most probably as a result of trea | atment for a previously existing ma | alignancy. | |
| Tumor pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder characterize | ed by marked discomfort from a ne | eoplasm that may be pressing on | a nerve, blocking blood vessels, ir | nflamed or fractured from metastas | sis. |
| Neoplasms benign, malignant<br>and unspecified (incl cysts and<br>polyps) - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Nervous system disorders | | | | |
|---|---|---|---|---|---|
| Grade | | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abducens nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | zed by involvement of the abducen | s nerve (sixth cranial nerve). | 1 | I | 1 |
| Accessory nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the accessor | ry nerve (eleventh cranial nerve). | | <b>-</b> | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by involvement of the acoustic | nerve (eighth cranial nerve). | | T | |
| Akathisia | Mild restlessness or increased motor activity | Moderate restlessness or increased motor activity; limiting instrumental ADL | Severe restlessness or increased motor activity; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by an uncomfortable feeling of | inner restlessness and inability to | stay still; this is a side effect of so | me psychotropic drugs. | |
| Amnesia | Mild; transient memory loss | Moderate; short term memory loss; limiting instrumental ADL | Severe; long term memory loss;<br>limiting self care ADL | - | - |
| | zed by systematic and extensive lo | ss or memory. | V-: | | T |
| Aphonia | - | - | Voicelessness; unable to speak | 1 | 1- |
| Definition: A disorder characteriz | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by inflammation of the arachno | id membrane and adjacent subara | achnoid space. | | |
| Ataxia | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; mechanical assistance indicated | - | - |
| Definition: A disorder characteriz | zed by lack of coordination of musc | ।<br>ale movements resulting in the imp | 1 | ı<br>ıntarv activities. | 1 |
| Brachial plexopathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz | zed by regional paresthesia of the l | brachial plexus, marked discomfor | t and muscle weakness, and limite | ed movement in the arm or hand. | |
| Central nervous system<br>necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms;<br>corticosteroids indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by a necrotic process occurring | in the brain and/or spinal cord. | 1 | I | , |
| Cerebrospinal fluid leakage | Post-craniotomy: asymptomatic;<br>Post-lumbar puncture: transient<br>headache; postural care<br>indicated | Post-craniotomy: moderate<br>symptoms; medical intervention<br>indicated; Post-lumbar<br>puncture: persistent moderate<br>symptoms; blood patch<br>indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | zed by loss of cerebrospinal fluid in | to the surrounding tissues. | T | T | |
| Cognitive disturbance | Mild cognitive disability; not<br>interfering with work/school/life<br>performance; specialized<br>educational services/devices<br>not indicated | Moderate cognitive disability;<br>interfering with work/school/life<br>performance but capable of<br>independent living; specialized<br>resources on part time basis<br>indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | - | - |
| Definition: A disorder characterize | zed by a conspicuous change in co | gnitive function. | 1 | T | |
| Concentration impairment | Mild inattention or decreased level of concentration | Moderate impairment in attention or decreased level of concentration; limiting instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | - | - |

| Nervous system disorders Grade | | | | | |
|---|---|---|---|---|---|
| Advance Event | 4 | | | 4 | |
| Adverse Event | Decrees distributed of slowly and | 2 | 3 | | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to stimuli; limiting instrumental ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder characte | rized by a decrease in ability to perc | eive and respond. | • | | |
| Dizziness | Mild unsteadiness or sensation | Moderate unsteadiness or | Severe unsteadiness or | - | - |
| | of movement | sensation of movement; limiting instrumental ADL | sensation of movement; limiting self care ADL | | |
| Definition: A disorder characte | rized by a disturbing sensation of lig | htheadedness, unsteadiness, gidd | liness, spinning or rocking. | | |
| Dysarthria | Mild slurred speech | Moderate impairment of articulation or slurred speech | Severe impairment of articulation or slurred speech | - | - |
| Definition: A disorder characte | rized by slow and slurred speech re | sulting from an inability to coordina | te the muscles used in speech. | · | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration;<br>limiting self care ADL | - | - |
| Definition: A disorder characte | rized by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation. | | |
| Dysgeusia | Altered taste but no change in diet | Altered taste with change in diet (e.g., oral supplements); noxious or unpleasant taste; loss of taste | - | - | - |
| Definition: A disorder characte | rized by abnormal sensual experien | ince with the taste of foodstuffs; it ca | n be related to a decrease in the s | sense of smell. | 1 |
| Dysphasia | Awareness of receptive or expressive characteristics; not impairing ability to communicate | Moderate receptive or expressive characteristics; impairing ability to communicate spontaneously | Severe receptive or expressive characteristics; impairing ability to read, write or communicate intelligibly | - | - |
| Definition: A disorder characte | rized by impairment of verbal comm | unication skills, often resulting fron | n brain damage. | <del></del> | 1 |
| Edema cerebral | - | - | - | Life-threatening consequences; urgent intervention indicated | - |
| Definition: A disorder characte | rized by swelling due to an excessiv | e accumulation of fluid in the brain | l. | Т | 1 |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a pathologic process involving | ng the brain. | 1 | Г | |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary<br>movements; limiting<br>instrumental ADL | Severe involuntary movements or torticollis; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by abnormal, repetitive, involu | ntary muscle movements, frenzied | speech and extreme restlessness | ·<br>S. | |
| Facial muscle weakness | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a reduction in the strength of | of the facial muscles. | | _ | |
| Facial nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by involvement of the facial ne | rve (seventh cranial nerve). | | | |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by involvement of the glossoph | naryngeal nerve (ninth cranial nerv | e). | | |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by a sensation of marked disco | omfort in various parts of the head | , not confined to the area of distrib | ution of any nerve. | |
| Hydrocephalus | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; intervention not indicated | Severe symptoms or neurological deficit; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal increase of ce | rebrospinal fluid in the ventricles o | f the brain. | ·<br> | |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | - | - |
| Deficition: A disconder observator | rized by characterized by excessive | | | • | • |

| Nervous system disorders | | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| | | | Grade | 1 | 1 | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 | | | |
| Hypoglossal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| Definition: A disorder characteriz | zed by involvement of the hypoglos | ssal nerve (twelfth cranial nerve). | • | • | | | | |
| Intracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death | | | |
| Definition: A disorder characteriz | zed by bleeding from the cranium. | | | | | | | |
| Ischemia cerebrovascular | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | - | - | - | | | |
| Definition: A disorder characteriz<br>damage. | zed by a decrease or absence of b | lood supply to the brain caused by | obstruction (thrombosis or embol | ism) of an artery resulting in neuro | ological | | | |
| IVth nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| Definition: A disorder characterize | zed by involvement of the trochlear | nerve (fourth cranial nerve). | I | T | | | | |
| Lethargy | Mild symptoms; reduced alertness and awareness | Moderate symptoms; limiting instrumental ADL | - | - | - | | | |
| Definition: A disorder characterization | zed by a decrease in consciousnes | s characterized by mental and ph | ysical inertness. | T | | | | |
| Leukoencephalopathy | Asymptomatic; small focal T2/FLAIR hyperintensities; involving periventricular white matter or <1/3 of susceptible areas of cerebrum +/- mild increase in subarachnoid space (SAS) and/or mild ventriculomegaly | Moderate symptoms; focal T2/FLAIR hyperintensities, involving periventricular white matter extending into centrum semiovale or involving 1/3 to 2/3 of susceptible areas of cerebrum +/- moderate increase in SAS and/or moderate ventriculomegaly | +/- moderate to severe increase | Life-threatening consequences; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly | Death | | | |
| Definition: A disorder characterize | '<br>zed by diffuse reactive astrocytosis | with multiple areas of necrotic for | i without inflammation. | ' | | | | |
| Memory impairment | Mild memory impairment | Moderate memory impairment; | Severe memory impairment;<br>limiting self care ADL | - | - | | | |
| Definition: A disorder characteriz | zed by a deterioration in memory fu | ınction. | | | | | | |
| Meningismus | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death | | | |
| Definition: A disorder characteriz | zed by neck stiffness, headache, a | nd photophobia resulting from irrit | ation of the cerebral meninges. | | | | | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| Definition: A disorder characteriz | zed by uncontrolled and purposeles | ss movements. | 1 | 1 | 1 | | | |
| Myelitis | Asymptomatic; mild signs (e.g.,<br>Babinski's reflex or Lhermitte's<br>sign) | Moderate weakness or sensory loss; limiting instrumental ADL | Severe weakness or sensory loss; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death | | | |
| Definition: A disorder characteriz | zed by inflammation involving the s | pinal cord. Symptoms include wea | akness, paresthesia, sensory loss, | marked discomfort and incontiner | nce. | | | |
| Neuralgia | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - | | | |
| Definition: A disorder characterize | zed by intense painful sensation alo | | I | I | | | | |
| Nystagmus | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| Definition: A disorder characterize | zed by involuntary movements of the | ne eyeballs. | I | T | | | | |
| Oculomotor nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| Definition: A disorder characteriz | zed by involvement of the oculomo | tor nerve (third cranial nerve). | 1 | 1 | | | | |
| Olfactory nerve disorder | - | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - | | | |
| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | · | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characteriz are experienced in the absence of | | ensory neurons resulting in abnor | mal cutaneous sensations of tinglin | ng, numbness, pressure, cold, and | warmth that |
| Peripheral motor neuropathy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneration | on of the peripheral motor nerves. | | | |
| Peripheral sensory neuropathy | Asymptomatic; loss of deep tendon reflexes or paresthesia | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | | on of the peripheral sensory nerve | | | |
| Phantom pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| | ed by marked discomfort related to | | ed from or is not physically part of | the body. | |
| Presyncope | - | Present (e.g., near fainting) | - | - | - |
| | | ess and dizziness which may prec | | | |
| Pyramidal tract syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ed by dysfunction of the corticospi<br>nd a decrease in fine motor coord | | l cord. Symptoms include an incre | ease in the muscle tone in the lowe | er extremities, |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting instrumental ADL; medical intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz connecting nerve root. | ed by inflammation involving a ne | rve root. Patients experience mark | ed discomfort radiating along a ne | erve path because of spinal pressu | re on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by paralysis of the recurrent la | ryngeal nerve. | | | |
| Reversible posterior leukoencephalopathy syndrome | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; abnormal imaging studies; limiting instrumental ADL | Severe symptoms; very<br>abnormal imaging studies;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | - | = | | findings of posterior leukoencepha<br>s an acute or subacute reversible o | |
| Seizure | Brief partial seizure; no loss of consciousness | Brief generalized seizure | Multiple seizures despite medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characteriz | ed by a sudden, involuntary skele | tal muscular contractions of cereb | ral or brain stem origin. | T | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteriz | ed by marked discomfort in the fac | ce, between the eyes, or upper tee | eth originating from the sinuses. | 1 | ı |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by characterized by excessive | sleepiness and drowsiness. | | | |
| Spasticity | Mild or slight increase in muscle tone | Moderate increase in muscle<br>tone and increase in resistance<br>through range of motion | Severe increase in muscle tone and increase in resistance through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characteriz disturbances. | ed by increased involuntary musc | | | It results in gait, movement, and s | peech |
| Stroke | Asymptomatic or mild neurologic deficit; radiographic findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a sudden loss of sensory fu | nction due to an intracranial vascu | ılar event. | 1 | ı |
| Syncope Definition: A disorder characteriz | -<br>ed by spontaneous loss of conscie | -<br>cusness caused by insufficient blo | Fainting; orthostatic collapse od supply to the brain. | - | - |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Transient ischemic attacks | Mild neurologic deficit with or without imaging confirmation | Moderate neurologic deficit with or without imaging confirmation | - | - | - |
| Definition: A disorder characterize | ed by a brief attack (less than 24 h | nours) of cerebral dysfunction of va | ascular origin, with no persistent n | eurological deficit. | |
| Tremor | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by the uncontrolled shaking mo | evement of the whole body or indiv | ridual parts. | | |
| Trigeminal nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by involvement of the trigemina | al nerve (fifth cranial nerve). | | | |
| Vagus nerve disorder | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by involvement of the vagus ne | rve (tenth cranial nerve). | • | | |
| Vasovagal reaction | - | - | Present | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize increase in the stimulation of the | ed by a sudden drop of the blood p | pressure, bradycardia, and periph | eral vasodilation that may lead to | loss of consciousness. It results fr | om an |
| Nervous system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Pregna | ancy, puerperium and pe | rinatal conditions | | |
|---|---|---|---|---|
| Grade | | | | |
| 1 | 2 | 3 | 4 | 5 |
| • | • | - | - | Fetal loss at<br>any<br>gestational<br>age |
| • | product of conception to show evi | dence of respiration, heartbeat, or | definite movement of a voluntary | muscle after |
| t possibility of resuscitation. | | | | |
| - | <10% percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | - |
| ed by inhibition of fetal growth resu | ulting in the inability of the fetus to | achieve its potential weight. | | |
| • | • | Delivery of a liveborn infant at 24 to 28 weeks gestation | Delivery of a liveborn infant at 24 weeks of gestation or less | - |
| ed by delivery of a viable infant be | fore the normal end of gestation. | Typically, viability is achievable be | tween the twentieth and thirty-sev | enth week of |
| - | - | Unintended pregnancy | - | - |
| ed by an unexpected pregnancy a | t the time of conception. | • | • | ' |
| • • | | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | ted by death in utero; failure of the t possibility of resuscitation. - ted by inhibition of fetal growth resurce downward of a liveborn infant at >34 to 37 weeks gestation and by delivery of a viable infant be ted by an unexpected pregnancy at Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention | ted by death in utero; failure of the product of conception to show evit possibility of resuscitation. - | The dead by death in utero; failure of the product of conception to show evidence of respiration, heartbeat, or to possibility of resuscitation. - | The dead by death in utero; failure of the product of conception to show evidence of respiration, heartbeat, or definite movement of a voluntary to possibility of resuscitation. - <10% percentile of weight for gestational age <5% percentile of weight for gestational age <1% percentile of weight for |

| | | Psychiatric disor | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation; hospitalization not indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by a state of restlessness asso | | irritability and tension. | | |
| Anorgasmia | Inability to achieve orgasm not adversely affecting relationship | Inability to achieve orgasm adversely affecting relationship | - | - | - |
| | erized by an inability to achieve orgas | | | | |
| Anxiety | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization not indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder characte stimulus. | erized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dys | pnea unattached to a clearly iden | tifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by a lack of clear and orderly the | nought and behavior. | | | |
| Delayed orgasm | | Delay in achieving orgasm adversely affecting relationship | - | - | - |
| | erized by sexual dysfunction characte | | T | I | I_ |
| Delirium | Mild acute confusional state | Moderate and acute confusional state; limiting instrumental ADL | Severe and acute confusional state; limiting self care ADL; hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder character reversible condition. | erized by the acute and sudden devel | opment of confusion, illusions, mo | ovement changes, inattentiveness, | agitation, and hallucinations. Usu | ally, it is a |
| Delusions | - | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by false personal beliefs held c | ontrary to reality, despite contradi | ctory evidence and common sense | e. | |
| Depression | Mild depressive symptoms | Moderate depressive symptoms; limiting instrumental ADL | Severe depressive symptoms;<br>limiting self care ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by melancholic feelings of grief | or unhappiness. | ' | ' | • |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | - |
| Definition: A disorder characte | erized by an exaggerated feeling of w | ell-being which is disproportionate | to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | Death |
| Definition: A disorder characte | erized by a false sensory perception i | n the absence of an external stimu | ılus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling asleep, staying asleep or waking up early | Severe difficulty in falling asleep, staying asleep or waking up early | - | - |
| Definition: A disorder characte | erized by difficulty in falling asleep an | d/or remaining asleep. | | | |
| Libido decreased | Decrease in sexual interest not adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | - | - | - |
| Definition: A disorder characte | erized by a decrease in sexual desire | T | 1 | T | 1 |
| Libido increased | Mild increase in sexual interest not adversely affecting relationship | Moderate increase in sexual interest adversely affecting relationship | Severe increase in sexual interest leading to dangerous behavior | - | - |
| Definition: A disorder characte | erized by an increase in sexual desire | ). | | | |
| Mania | Mild manic symptoms (e.g.,<br>elevated mood, rapid thoughts,<br>rapid speech, decreased need<br>for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characte | erized by excitement of psychotic prop | oortions manifested by mental and | l physical hyperactivity, disorganiz | ation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |

| | | Psychiatric disord | ders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterize | ed by a conspicuous change in a p | person's behavior and thinking. | | | |
| Psychosis | Mild psychotic symptoms | Moderate psychotic symptoms<br>(e.g., disorganized speech;<br>impaired reality testing) | Severe psychotic symptoms<br>(e.g., paranoid; extreme<br>disorganization); hospitalization<br>not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder characterize tumor. | ed by personality change, impaired | d functioning, and loss of touch wi | th reality. It may be a manifestatio | n of schizophrenia, bipolar disorde | er or brain |
| Restlessness | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by an inability to rest, relax or b | e still. | | | |
| Suicidal ideation | Increased thoughts of death but no wish to kill oneself | Suicidal ideation with no specific plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide<br>with serious intent to die which<br>requires hospitalization | - |
| Definition: A disorder characterize | ed by thoughts of taking one's owr | n life. | | | |
| Suicide attempt | - | - | Suicide attempt or gesture without intent to die which may not require hospitalization | Suicide attempt with intent to die which requires hospitalization | Death |
| Definition: A disorder characterize | ed by self-inflicted harm in an atter | mpt to end one's own life. | | | |
| Psychiatric disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting<br>self care ADL | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |

| | | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Acute kidney injury | Creatinine level increase of >0.3 mg/dL; creatinine 1.5 - 2.0 x above baseline | baseline | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated | Life-threatening consequences; dialysis indicated | Death |
| Definition: A disorder character<br>causes (ureteral or bladder out | rized by the acute loss of renal functi<br>flow obstruction). | ion and is traditionally classified a | s pre-renal (low blood flow into kid | ney), renal (kidney damage) and բ | oost-renal |
| Bladder perforation | - | Extraperitoneal perforation, indwelling catheter indicated | Intraperitoneal perforation;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by a rupture in the bladder wall | | | | |
| Bladder spasm | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | - | - |
| Definition: A disorder character | rized by a sudden and involuntary co | ontraction of the bladder wall. | | • | |
| Chronic kidney disease | eGFR (estimated Glomerular<br>Filtration Rate) or CrCl<br>(creatinine clearance) <lln -="" 60<br="">ml/min/1.73 m2 or proteinuria<br/>2+ present; urine<br/>protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl <15 ml/min/1.73<br>m2; dialysis or renal transplant<br>indicated | Death |
| Definition: A disorder character | ized by gradual and usually perman | ent loss of kidney function resultir | ng in renal failure. | | |
| Cystitis noninfective | Microscopic hematuria; minimal increase in frequency, urgency, dysuria, or nocturia; new onset of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the bladder | ,<br>which is not caused by an infection | on of the urinary tract. | • | • |
| Hematuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; urinary catheter or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV medications or hospitalization indicated; elective endoscopic, radiologic or operative intervention indicated; limiting self care ADL | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder character | rized by laboratory test results that in | ndicate blood in the urine. | | T | |
| Hemoglobinuria | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate the presence of free hemo | oglobin in the urine. | | |
| Proteinuria | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs | Adults: 2+ proteinuria; urinary<br>protein 1.0 - 3.4 g/24 hrs;<br>Pediatric: urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5<br>g/24 hrs;<br>Pediatric: urine P/C >1.9 | - | - |
| Definition: A disorder character | ized by laboratory test results that ir | ndicate the presence of excessive | protein in the urine. It is predomin | antly albumin, but also globulin. | |
| Renal calculi | Asymptomatic or mild symptoms; occasional use of nonprescription analgesics indicated | Symptomatic; oral antiemetics indicated; around the clock nonprescription analgesics or any oral narcotic analgesics indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences;<br>urgent radiologic, endoscopic or<br>operative intervention indicated | Death |
| Definition: A disorder character | rized by the formation of crystals in t | he pelvis of the kidney. | T | T | |
| Renal colic | Mild pain not interfering with activity; nonprescription medication indicated | Moderate pain; limiting instrumental ADL; prescription medication indicated | Hospitalization indicated;<br>limiting self care ADL | - | - |

| | | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or<br>hospitalization indicated;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the kidney. | | | | |
| Urinary fistula | - | Noninvasive intervention indicated; urinary or suprapubic catheter placement indicated | Limiting self care ADL; elective<br>radiologic, endoscopic or<br>operative intervention indicated;<br>permanent urinary diversion<br>indicated | Life-threatening consequences; urgent radiologic or operative intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between any part of the urinary s | system and another organ or anato | omic site. | |
| Urinary frequency | Present | Limiting instrumental ADL; medical management indicated | - | - | - |
| Definition: A disorder characteri | zed by urination at short intervals. | Т | T | Т | 1 |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>limiting instrumental ADL | Intervention indicated (e.g., clamp, collagen injections); operative intervention indicated; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by inability to control the flow o | f urine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or intermittent catheter placement not indicated; able to void with some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Life-threatening consequences; organ failure; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by accumulation of urine within | the bladder because of the inabil | ity to urinate. | | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by blockage of the normal flow | of contents of the urinary tract. | T | T | 1 |
| Urinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the urinary tract. | 1 | T | |
| Urinary urgency | Present | Limiting instrumental ADL;<br>medical management indicated | - | - | - |
| Definition: A disorder characteri | zed by a sudden compelling urge to | o urinate. | T | T | 1 |
| Urine discoloration | Present | - | - | - | - |
| Definition: A disorder characteri | zed by a change in the color of the | urine. | 1 | T | |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azoospermia | - | - | Absence of sperm in ejaculate | - | - |
| Definition: A disorder characte | erized by laboratory test results that ir | ndicate complete absence of speri | matozoa in the semen. | | • |
| Breast atrophy | Minimal asymmetry; minimal | Moderate asymmetry; moderate | Asymmetry >1/3 of breast | - | - |
| | atrophy | atrophy | volume; severe atrophy | | |
| Definition: A disorder characte | erized by underdevelopment of the br | east. | | | , |
| Breast pain | Mild pain | Moderate pain; limiting | Severe pain; limiting self care | - | _ |
| | · | instrumental ADL | ADL | | |
| Definition: A disorder characte | erized by marked discomfort sensation | n in the breast region. | ' | • | • |
| Dysmenorrhea | Mild symptoms; intervention not | | Severe symptoms; limiting self | _ | _ |
| -, | indicated | instrumental ADL | care ADL | | |
| Definition: A disorder characte | erized by abnormally painful abdomina | al cramps during menses. | ! | ! | ' |
| Dyspareunia | Mild discomfort or pain | Moderate discomfort or pain | Severe discomfort or pain | | |
| Jyspareuma | associated with vaginal | associated with vaginal | associated with vaginal | - | - |
| | penetration; discomfort relieved | penetration; discomfort or pain | penetration; discomfort or pain | | |
| | with use of vaginal lubricants or | partially relieved with use of | unrelieved by vaginal lubricants | | |
| | estrogen | vaginal lubricants or estrogen | or estrogen | | |
| Definition: A disorder characte | erized by painful or difficult coitus. | • | | | , |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde | _ | _ | - |
| | Januario ejasanansi. | ejaculation | | | |
| Definition: A disorder characte | rized by problems related to ejaculat | 1 - | ı<br>ture, delayed, retrograde and pair | ı<br>ıful ejaculation | 1 |
| Erectile dysfunction | Decrease in erectile function | Decrease in erectile function | Decrease in erectile function | liui ojuoululion. | |
| Erectile dystatiction | (frequency or rigidity of | (frequency/rigidity of erections), | (frequency/rigidity of erections) | - | - |
| | erections) but intervention not | erectile intervention indicated, | but erectile intervention not | | |
| | indicated (e.g., medication or | (e.g., medication or mechanical | helpful (e.g., medication or | | |
| | use of mechanical device, | devices such as penile pump) | mechanical devices such as | | |
| | penile pump) | | penile pump); placement of a | | |
| | | | permanent penile prosthesis | | |
| | | | indicated (not previously | | |
| | | | present) | | |
| Definition: A disorder characte | erized by the persistent or recurrent in | nability to achieve or to maintain a | n erection during sexual activity. | | |
| Fallopian tube obstruction | Diagnostic observations only; | Mild symptoms; elective | Severe symptoms; elective | - | - |
| · | intervention not indicated | intervention indicated | operative intervention indicated | | |
| Definition: A disorder characte | erized by blockage of the normal flow | of the contents in the fallopian tub | pe. | ' | • |
| Fallopian tube stenosis | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| anopian tago otonosio | diagnostic observations only; | not indicated | operative intervention indicated | urgent operative intervention | J Suil. |
| | intervention not indicated | | ' | indicated (e.g., organ resection) | |
| Definition: A disorder characte | erized by a narrowing of the fallopian | r<br>tube lumen | ı | | ' |
| Female genital tract fistula | Asymptomatic clinical or | Symptomatic and intervention | Severe symptoms; elective | Life-threatening consequences; | Death |
| i emale gemilai traci nstula | diagnostic observations only; | not indicated | operative intervention indicated | urgent intervention indicated | Death |
| | intervention not indicated | The maiotica | operative intervention interest | angone micromicon maioatou | |
| Definition: A disorder characte | ा<br>erized by an abnormal communicatior | l<br>n hetween a female renroductive s | l<br>system organ and another organ o | r anatomic site | 1 |
| | | | ystem organ and another organ o | anatomic site. | 1 |
| Feminization acquired | Mild symptoms; intervention not indicated | intervention indicated | - | - | - |
| D-fi-iti A didb | ı | 1 | | l | I |
| | erized by the development of secondar | l' | | | |
| Genital edema | Mild swelling or obscuration of | Readily apparent obscuration of | Lymphorrhea; gross deviation | - | - |
| | anatomic architecture on close | anatomic architecture; | from normal anatomic contour; | | |
| | inspection | obliteration of skin folds; readily | limiting self care ADL | | |
| | | apparent deviation from normal anatomic contour | | | |
| Definition: A disorder characte | I<br>arized by swelling due to an excessive | ı | l<br>ale | I | I |
| | erized by swelling due to an excessive | | | | |
| Gynecomastia | Asymptomatic breast | Symptomatic (e.g., pain or | Severe symptoms; elective | - | - |
| | enlargement | psychosocial impact) | operative intervention indicated | I | I |
| Definition: A disorder characte | erized by excessive development of the | ne breasts in males. | T | T | |
| Hematosalpinx | Minimal bleeding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| | imaging study or laparoscopy; | intervention indicated | indicated; radiologic or | urgent operative intervention | |
| | intervention not indicated | | endoscopic intervention | indicated | |
| | | i . | indicated | | |

| Adverse Event 1 2 9 9 9 9 9 9 9 9 9 9 9 9 9 9 9 9 9 9 | |
|---|---|
| Definition: A disorder characterized by the presence of blood in a failopian tube. Intermittent menses with along the minimal bleam infermittent menses with along the menses for more than 1 to 3 months along the menses for more than 1 to 3 months. Befinition: A disorder characterized by tragular cycle or duration of menses. Lactation disorder Mid changes in lactation, not aganificantly affecting production or expression of breast misk. Definition: A disorder characterized by disturbances of milk secretion. It is not necessarily related to pregnancy that is observed in females and can be observed from the control of the production or expression of breast misk. Definition: A disorder characterized by abnormally heavy varginal bleeding during menses. Nippilo deformity Asymptomatic, asymmetry with alight retraction and/or thickening of the nippile aerodar complex or complex. Symptomatic, asymmetry of thickening of the nippile aerodar complex with moderate treation and/or thickening of the nippile aerodar complex with moderate treation and/or thickening of the nippile aerodar complex with moderate treation and/or indicated (as graph of the nippile aerodar complex with moderate treation and/or indicated by a decrease in the number of spentrum or moderated by a decrease in the number of spentrum or moderated and the number of spentrum or moderated in the number of spentrum or moderated and the number of spentrum or moder | |
| Intermittent menses with aksped menses (or no more laksped menses (or no more laksped menses for more laksped menses for no menses. Lactation disorder characterized by a disturbance of milk penses for no more laksped menses for no more laksped menses for no more laksped menses for no menses. Definition: A disorder characterized by a malformation of the nipple areadar complex with hickening of the nipple areadar complex with hickening of the nipple areadar complex with hickening of the nipple areadar complex with hickening of the nipple areadar consists of the number of sperme concentration 13 - 48 million/mil. or motility 2-52 Million/million: A disorder char | 5 |
| befinition: A disorder characterized by disturbances of milk secretion. It is not necessarily related to pregular cycle or duration of membes. Lectation disorder Mild changes in lactation, not significantly affecting production or expression of breast milk or expression or breast milk or expression or b | |
| Lactation disorder Mild changes in lactation, not significantly affecting production of repression of breast milk production or expression or production or expression or production or production or expression or production or expression or production or expression or production or expression or production or produ | - |
| significantly affecting production or expression of breast milk and production or expression or production or expression and production or expression or production or expression or production or expression or production or expression or production or | |
| Memorrhagia | - |
| Intervention indicated (e.g., hysterectomy) Intervention indicated (e.g., hysterectomy) | d in males. |
| Asymptomatic; asymmetry with slight retraction and/or thickening of the nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex Definition: A disorder characterized by a maiformation of the nipple. Oligospermia Sperm concentration >48 million/mL or motility >68% million/mL or motility <52% Definition: A disorder characterized by the deeding identified on imaging study or laproscopy; intervention not indicated with revention pain with dispain with revention in one side of the abdomen between menstrual cycles, around the time of the discharge of ovarian folicle. Definition: A disorder characterized by marked discomfort sensation in one side of the abdomen between menstrual cycles, around the time of the discharge of ovarian folicle. Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Definition: A disorder characterized by marked discomfort sensation in the pelvis. Definition: A disorder characterized by marked discomfort sensation in the pelvis. Definition: A disorder characterized by marked discomfort se | |
| slight retraction and/or thickening of the nipple areolar complex with moderate retraction and/or thickening of the nipple areolar complex complex Definition: A disorder characterized by a maiformation of the nipple. Digospermia Sperm concentration >48 million/mL or motility >68% million/mL or motility >68% million/mL or motility >32 - 68% million/mL or motil | |
| Sperm concentration > 48 million/mL or motility > 68% million/mL or motility > 32 - 68% million/mL or moti | - |
| Definition: A disorder characterized by a decrease in the number of spermatozoa in the semen. Ovarian hemorrhage | |
| Minimal bleeding identified on imaging study or laproscopy; intervention not indicated Definition: A disorder characterized by bleeding from the ovary. Ovarian rupture Asymptomatic clinical or diagnostic observations only; intervention of the ovarian stibution pain Mild pain Moderate plan; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mid pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mid pain Moderate pain; limiting instrumental ADL Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Life-threatening conse urgent intervention indicated urgent intervention indicated urgent intervention indicated instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mid pain Moderate pain; limiting severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mid pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mid pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. | - |
| imaging study or laproscopy; intervention not indicated Definition: A disorder characterized by bleeding from the ovary. Ovarian rupture Asymptomatic clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by tearing or disruption of the ovarian tissue. Ovulation pain Mild pain Moderate pain; limiting intervention Moderate pain; limiting intervention Moderate pain; limiting intervention Moderate pain; limiting intervention Moderate pain; limiting intervention Moderate pain; limiting Severe symptoms; limiting self care diagnostic observations only; intervention indicated Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting Severe pain; limiting self care aDL Life-threatening conse urgent intervention indi Life-threatening conse urgent intervention ind Life-threatening conse urgent intervention ind Life-threatening conse urgent intervention ind Life-threatening conse urgent intervention ind Life-threatening conse urgent intervention ind Severe symptoms; limiting self care ADL Life-threatening conse urgent intervention ind Moderate pain; limiting intervention ind Severe pain; limiting self care ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting instrumental ADL ADL Definition: A disorder characterized by marked discomfort sensation in the peris. Perineal pain Moderate pain; limiting instrumental ADL ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | |
| Asymptomatic clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by tearing or disruption of the ovariant tissue. Doulation pain Mild pain Moderate pain; limiting sever pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in one side of the abdomen between menstrual cycles, around the time of the discharge of diagnostic observations only; intervention not indicated Definition: A disorder characterized by marked discomfort sensation in one side of the abdomen between menstrual cycles, around the time of the discharge of diagnostic observations only; intervention not indicated Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Penile pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | |
| diagnostic observations only; intervention not indicated Definition: A disorder characterized by tearing or disruption of the ovarian tissue. Ovulation pain Mid pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by marked discomfort sensation in one side of the abdomen between menstrual cycles, around the time of the discharge of diagnostic observations only; intervention not indicated Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mid pain Moderate pain; limiting Severe pain; limiting self care ADL Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mid pain Moderate pain; limiting Initing Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mid pain Moderate pain; limiting Initing Init | ' |
| Ovulation pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by marked discomfort sensation in one side of the abdomen between menstrual cycles, around the time of the discharge covarian follicle. Pelvic floor muscle weakness Asymptomatic; clinical or diagnostic observations only; intervention not indicated Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting seven menstrual cycles, around the time of the discharge of the discharge of the pelvic floor. Symptomatic, not interfering with bladder, bowel, or vaginal function; limiting instrumental ADL ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pa | |
| instrumental ADL ADL Definition: A disorder characterized by marked discomfort sensation in one side of the abdomen between menstrual cycles, around the time of the discharge of covarian follicle. Pelvic floor muscle weakness Asymptomatic; clinical or diagnostic observations only; intervention not indicated intervention not indicated with bladder, bowel, or vaginal function; limiting instrumental ADL Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | ' |
| Ovarian follicle. Pelvic floor muscle weakness | - |
| diagnostic observations only; intervention not indicated six of the pelvic floor. Definition: A disorder characterized by a reduction in the strength of the muscles of the pelvic floor. Pelvic pain Mild pain Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting instrumental ADL ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting instrumental ADL ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | f the ovum from the |
| Pelvic pain Mild pain Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | |
| instrumental ADL Definition: A disorder characterized by marked discomfort sensation in the pelvis. Penile pain Mild pain Moderate pain; limiting instrumental ADL ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting instrumental ADL Moderate pain; limiting instrumental ADL Severe pain; limiting instrumental ADL ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | |
| Penile pain Mild pain Moderate pain; limiting instrumental ADL Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting self care and pain; limiting instrumental ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | - |
| instrumental ADL ADL Definition: A disorder characterized by marked discomfort sensation in the penis. Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care instrumental ADL ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | |
| Perineal pain Mild pain Moderate pain; limiting Severe pain; limiting self care - ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | - |
| instrumental ADL ADL Definition: A disorder characterized by a sensation of marked discomfort in the area between the genital organs and the anus. | <del></del> |
| | - |
| Premature menopause - - Present - | |
| | - |
| Definition: A disorder characterized by ovarian failure before the age of 40. Symptoms include hot flashes, night sweats, mood swings and a decrease in sex of the following states of the flashes and the flashes, night sweats, mood swings and a decrease in sex of the flashes, mood swings and a decrease in sex of the flashes, mood swings and a decrease in sex of the flashes, mood swings and a decrease in sex of the flashes, mood swings and a decrease in sex of the flashes, mood swings and a decrease in sex | quences; Death |

| Reproductive system and breast disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | 1 |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characterized | zed by bleeding from the prostate of | gland. | 1 | | |
| Prostatic obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| | zed by compression of the urethra | secondary to enlargement of the p | prostate gland. This results in voidi | ng difficulties (straining to void, slo | ow urine |
| stream, and incomplete emptyin | · | T | T | | 1 |
| Prostatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the prostate gland. | | | |
| Scrotal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensatio | n in the scrotal area. | | | |
| Spermatic cord hemorrhage | Minimal bleeding identified on imaging study; intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characteri | zed by bleeding from the spermatic | cord. | | | |
| Spermatic cord obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by blockage of the normal flow | of the contents of the spermatic c | 1 - | • | • |
| Testicular disorder | Asymptomatic; clinical or | Symptomatic but not interfering | Severe symptoms; interfering | Life-threatening consequences; | Death |
| | diagnostic observations only; | with urination or sexual | with urination or sexual function; | urgent intervention indicated | |
| | intervention not indicated | activities; intervention not indicated; limiting instrumental ADL | limiting self care ADL;<br>intervention indicated | | |
| D-6:-:4: A did | | IVDE | l | | l |
| | zed by involvement of the testis. | | 0 11 5 4 6 5 | 126 11 1 1 | l |
| Testicular hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characterize | zed by bleeding from the testis. | | | | |
| Testicular pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by a sensation of marked disco | omfort in the testis. | ' | • | ' |
| Uterine fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between the uterus and another | organ or anatomic site. | ! | ' |
| | Minimal blooding identified on | Moderate bleeding; medical | Severe bleeding; transfusion | Life-threatening consequences; | Death |
| Uterine hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | intervention indicated | indicated; radiologic or<br>endoscopic intervention<br>indicated | urgent operative intervention indicated | |
| Ü | imaging study; intervention not indicated | | endoscopic intervention | | |
| Ü | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; | | endoscopic intervention indicated Severe symptoms; elective | | - |
| Definition: A disorder characteri.<br>Uterine obstruction | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; intervention not indicated | intervention indicated Mild symptoms; elective intervention indicated | endoscopic intervention indicated | | - |
| Definition: A disorder characteri:<br>Uterine obstruction<br>Definition: A disorder characteri: | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; | intervention indicated Mild symptoms; elective intervention indicated et. Moderate pain; limiting | endoscopic intervention indicated Severe symptoms; elective operative intervention indicated Severe pain; limiting self care | | - |
| Definition: A disorder characteri:<br>Uterine obstruction<br>Definition: A disorder characteri:<br>Uterine pain | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; intervention not indicated zed by blockage of the uterine outle Mild pain | intervention indicated Mild symptoms; elective intervention indicated et. Moderate pain; limiting instrumental ADL | endoscopic intervention indicated Severe symptoms; elective operative intervention indicated | | - |
| Definition: A disorder characteri: Uterine obstruction Definition: A disorder characteri: Uterine pain Definition: A disorder characteri: | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; intervention not indicated zed by blockage of the uterine outle Mild pain | mild symptoms; elective intervention indicated et. Moderate pain; limiting instrumental ADL comfort in the uterus. | endoscopic intervention indicated Severe symptoms; elective operative intervention indicated Severe pain; limiting self care | | - |
| Definition: A disorder characteri:<br>Uterine obstruction<br>Definition: A disorder characteri:<br>Uterine pain | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; intervention not indicated zed by blockage of the uterine outle Mild pain | intervention indicated Mild symptoms; elective intervention indicated et. Moderate pain; limiting instrumental ADL | endoscopic intervention indicated Severe symptoms; elective operative intervention indicated Severe pain; limiting self care | | - |
| Definition: A disorder characteri: Uterine obstruction Definition: A disorder characteri: Uterine pain Definition: A disorder characteri: Vaginal discharge | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; intervention not indicated zed by blockage of the uterine outled will pain zed by a sensation of marked disco | mild symptoms; elective intervention indicated et. Moderate pain; limiting instrumental ADL perfort in the uterus. Moderate to heavy vaginal discharge; use of perineal pad or tampon indicated | endoscopic intervention indicated Severe symptoms; elective operative intervention indicated Severe pain; limiting self care ADL | indicated - | |
| Definition: A disorder characteri: Uterine obstruction Definition: A disorder characteri: Uterine pain Definition: A disorder characteri: Vaginal discharge | imaging study; intervention not indicated zed by bleeding from the uterus. Diagnostic observations only; intervention not indicated zed by blockage of the uterine outle Mild pain zed by a sensation of marked discount | mild symptoms; elective intervention indicated et. Moderate pain; limiting instrumental ADL perfort in the uterus. Moderate to heavy vaginal discharge; use of perineal pad or tampon indicated | endoscopic intervention indicated Severe symptoms; elective operative intervention indicated Severe pain; limiting self care ADL | indicated - | ring years |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by an abnormal communication | between the vagina and another | organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on<br>clinical exam or imaging study;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion indicated; radiologic or endoscopic intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder characterize | ed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema, or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal ulceration; life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ed by inflammation involving the v | agina. Symptoms may include red | lness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only; intervention not indicated | Mild symptoms; elective intervention indicated | Severe symptoms; elective operative intervention indicated | - | - |
| Definition: A disorder characterize | ed by blockage of vaginal canal. | | 1 | 1 | |
| Vaginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characterize | ed by a sensation of marked disco | mfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or diagnostic observations only; intervention not indicated | Symptomatic and intervention not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characterize | ·<br>ed by a rupture in the vaginal wall. | | • | • | • |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or shortening not interfering with physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characterize | ed by a narrowing of the vaginal c | anal. | | | _ |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spasm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | - | - |
| Definition: A disorder characterize intercourse. | ed by involuntary spasms of the po | elvic floor muscles, resulting in pa | thologic tightness of the vaginal w | all during penetration such as duri | ng sexual |
| Reproductive system and breast disorders - Other, specify | * ' | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Adult respiratory distress<br>syndrome | - | - | Present with radiologic findings; intubation not indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri<br>surgery. | zed by progressive and life-threater | ning pulmonary distress in the abs | ence of an underlying pulmonary | condition, usually following major t | rauma or |
| Allergic rhinitis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| | zed by an inflammation of the nasa<br>s of the sinuses, eyes, middle ear, a | • | • | • | ay also |
| Apnea | - | - | Present; medical intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by cessation of breathing. | T | I | T | |
| Aspiration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Altered eating habits; coughing or choking episodes after eating or swallowing; medical intervention indicated (e.g., suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by inhalation of solids or liquids | s into the lungs. | | <u> </u> | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by the collapse of part or the en | ntire lung. | T | T | 1 |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | · | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., mild<br>wheezing); endoscopic<br>evaluation indicated;<br>radiographic evidence of<br>atelectasis/lobar collapse;<br>medical management indicated<br>(e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | zed by blockage of a bronchus pas | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor;<br>endoscopic intervention<br>indicated (e.g., laser, stent<br>placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | zed by a narrowing of the bronchial | 1 | | leg at the | <b>.</b> |
| Bronchopleural fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteri | zed by an abnormal communication | n between a bronchus and the ple | ural cavity. | I | |
| Bronchopulmonary hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g., | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention | Death |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | T | Grade | T | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Bronchospasm | Mild symptoms; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Limiting self care ADL; oxygen saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | rized by a sudden contraction of the | smooth muscles of the bronchial | wall. | | |
| Chylothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; thoracentesis or tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characte | rized by milky pleural effusion (abno | rmal collection of fluid) resulting fr | om accumulation of lymph fluid in | the pleural cavity. | |
| Cough | Mild symptoms; nonprescription intervention indicated | Moderate symptoms, medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte by a distinctive sound. | rized by sudden, often repetitive, spa | asmodic contraction of the thoraci | c cavity, resulting in violent release | e of air from the lungs and usually | accompani |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with minimal exertion; limiting instrumental ADL | Shortness of breath at rest;<br>limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an uncomfortable sensation | of difficulty breathing. | | | |
| Epistaxis | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated (e.g., nasal packing, cauterization; topical vasoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by bleeding from the nose. | 1 | 1 | 1 | |
| Hiccups | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe symptoms; interfering with sleep; limiting self care ADL | - | - |
| Definition: A disorder characte | rized by repeated gulp sounds that re | esult from an involuntary opening | and closing of the glottis. This is a | ttributed to a spasm of the diaphra | gm. |
| Hoarseness | Mild or intermittent voice change; fully understandable; self-resolves | Moderate or persistent voice<br>changes; may require<br>occasional repetition but<br>understandable on telephone;<br>medical evaluation indicated | Severe voice changes including predominantly whispered speech | - | - |
| Definition: A disorder characte | rized by harsh and raspy voice arisir | ng from or spreading to the larynx. | | | |
| Нурохіа | - | Decreased oxygen saturation<br>with exercise (e.g., pulse<br>oximeter <88%); intermittent<br>supplemental oxygen | Decreased oxygen saturation at<br>rest (e.g., pulse oximeter <88%<br>or PaO2 <=55 mm Hg) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | rized by a decrease in the level of ox | | 1. | l . | |
| Laryngeal edema | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | Stridor; respiratory distress;<br>hospitalization indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | rized by swelling due to an excessive | | | Ī | |
| _aryngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characte | ा<br>rized by an abnormal communication | between the larynx and another | organ or anatomic site. | , , | 1 |
| aryngeal hemorrhage | Mild cough or trace hemoptysis;<br>laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g., | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| | | | hemostasis of bleeding site) | Intabation) | ! |
| Definition: A disorder characte | rized by bleeding from the larynx. | | memostasis of bleeding site) | Intubation) | |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngeal mucositis | Endoscopic findings only; mild discomfort with normal intake | Moderate discomfort; altered oral intake | Severe pain; severely altered<br>eating/swallowing; medical<br>intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder characteri | ized by an inflammation involving th | e mucous membrane of the laryn | ζ. | İ | |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ized by blockage of the laryngeal ai | rway. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences; urgent intervention indicated | Death |
| | ized by a narrowing of the laryngea | | | | I |
| Laryngopharyngeal dysesthesia | a Mild symptoms; no anxiety;<br>intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspnea and swallowing difficulty; limiting self care ADL | Life-threatening consequences | Death |
| Definition: A disorder characteri | ized by an uncomfortable persistent | sensation in the area of the laryn | gopharynx. | | |
| Laryngospasm | - | Transient episode; intervention not indicated | Recurrent episodes;<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| Definition: A disorder characteri | ized by paroxysmal spasmodic mus | cular contraction of the vocal cord | | , , | 1 |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hemostasis of bleeding<br>site) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ा<br>ized by bleeding from the mediastin | um. | 1 / | l | 1 |
| Nasal congestion | Mild symptoms; intervention not indicated | | Associated with bloody nasal discharge or epistaxis | - | - |
| | ized by obstruction of the nasal pas | 1 | I | | 1 |
| Pharyngeal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | ized by an abnormal communication | n between the pharynx and anothe | er organ or anatomic site. | 1 | |
| Pharyngeal hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteri | ized by bleeding from the pharynx. | T | Т | Г | 1 |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics indicated; altered oral intake; limiting instrumental ADL | Severe pain; unable to<br>adequately aliment or hydrate<br>orally; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by an inflammation involving th | e mucous membrane of the phary | | | ı |
| Pharyngeal necrosis | - | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | Respir | ratory, thoracic and med | lastinal disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | rized by a necrotic process occurring | in the pharynx. | 1 | 1 | |
| Pharyngeal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder character | rized by a narrowing of the pharynge | al airway. | ' | ' | ' |
| Pharyngolaryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | - | - |
| Definition: A disorder character | rized by marked discomfort sensation | n in the pharyngolaryngeal region. | | <u> </u> | ı |
| Pleural effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., diuretics or limited therapeutic thoracentesis) | Symptomatic with respiratory<br>distress and hypoxia; surgical<br>intervention including chest tube<br>or pleurodesis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | rized by an increase in amounts of flo | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomfo | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage confirmed by thoracentesis | Symptomatic or associated with pneumothorax; chest tube drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder character | rized by bleeding from the pleural ca | vity. | • | • | • |
| Pleuritic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | rized by marked discomfort sensation | n in the pleura. | T | T | |
| Pneumonitis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL; oxygen indicated | Life-threatening respiratory compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | rized by inflammation focally or diffus | | | | I |
| Pneumothorax | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; intervention indicated (e.g., tube placement without sclerosis) | Sclerosis and/or operative intervention indicated; hospitalization indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by abnormal presence of air in | the pleural cavity resulting in the | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder character | rized by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | |
| Productive cough | | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | - | - |
| | rized by expectorated secretions upo | | Covere diannes er diannes et | Life threatening requireten. | Dooth |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at rest; oxygen indicated; limiting self care ADL | Life-threatening respiratory<br>compromise; urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder character | rized by accumulation of fluid in the I | | nce of the gas exchange that may | lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia; radiologic<br>pulmonary fibrosis <25% of lung<br>volume | Moderate hypoxemia; evidence<br>of pulmonary hypertension;<br>radiographic pulmonary fibrosis<br>25 - 50% | Severe hypoxemia; evidence of right-sided heart failure; radiographic pulmonary fibrosis >50 - 75% | Life-threatening consequences (e.g., hemodynamic/pulmonary complications); intubation with ventilatory support indicated; radiographic pulmonary fibrosis >75% with severe honeycombing | Death |
| Definition: A disorder character | rized by the replacement of the lung | tissue by connective tissue, leadir | ng to progressive dyspnea, respira | tory failure or right heart failure. | |
| Pulmonary fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL;<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |

| Respiratory, thoracic and mediastinal disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characteriz | red by an abnormal communication | between the lung and another or | gan or anatomic site. | <u> </u> | |
| Pulmonary hypertension | Minimal dyspnea; findings on physical exam or other evaluation | Moderate dyspnea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated<br>with hypoxemia, right heart<br>failure; oxygen indicated | Life-threatening airway<br>consequences; urgent<br>intervention indicated (e.g.,<br>tracheotomy or intubation) | Death |
| Definition: A disorder characteriz | ed by an increase in pressure with | in the pulmonary circulation due to | lung or heart disorder. | | |
| Respiratory failure | - | - | - | Life-threatening consequences; urgent intervention, intubation, or ventilatory support indicated | Death |
| Definition: A disorder characteriz<br>with an increase in arterial levels | red by impaired gas exchange by t<br>s of carbon dioxide. | he respiratory system resulting in | hypoxemia and a decrease in oxy | genation of the tissues that may be | e associate |
| Retinoic acid syndrome | Fluid retention; <3 kg of weight<br>gain; intervention with fluid<br>restriction and/or diuretics<br>indicated | Moderate signs or symptoms; steroids indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences; ventilatory support indicated | Death |
| Definition: A disorder characteriz retinoic acid. | zed by weight gain, dyspnea, pleur | al and pericardial effusions, leukoo | cytosis and/or renal failure original | ly described in patients treated wit | h all-trans |
| Sinus disorder | Asymptomatic mucosal crusting; blood-tinged secretions | Symptomatic stenosis or<br>edema/narrowing interfering<br>with airflow; limiting instrumental<br>ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone; urgent operative intervention indicated | Death |
| Definition: A disorder characteriz | red by involvement of the paranasa | al sinuses. | • | | |
| Sleep apnea | Snoring and nocturnal sleep arousal without apneic periods | Moderate apnea and oxygen<br>desaturation; excessive daytime<br>sleepiness; medical evaluation<br>indicated; limiting instrumental<br>ADL | Oxygen desaturation;<br>associated with hypertension;<br>medical intervention indicated;<br>limiting self care ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | red by cessation of breathing for sh | nort periods during sleep. | • | ' | • |
| Sneezing | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | - | - | - |
| Definition: A disorder characteriz | ed by the involuntary expulsion of | air from the nose. | | ' | ' |
| Sore throat | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | - | - |
| Definition: A disorder characteriz | red by of marked discomfort in the | throat | • | | |
| Stridor | - | - | Respiratory distress limiting self care ADL; medical intervention indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder characteriz | red by a high pitched breathing sou | und due to laryngeal or upper airw | ay obstruction. | | |
| Tracheal fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the trachea and another | organ or anatomic site. | | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe pain; hemorrhage or respiratory symptoms; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| | ted by an inflammation involving th | | | I | I_ |
| Tracheal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Stridor or respiratory distress<br>limiting self care ADL;<br>endoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| | red by a narrowing of the trachea. | 1 | • | • | • |

| | Respi | ratory, thoracic and med | iastinal disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Voice alteration | Mild or intermittent change from normal voice | Moderate or persistent change<br>from normal voice; still<br>understandable | Severe voice changes including predominantly whispered speech; may require frequent repetition or face-to-face contact for understandability; may require assistive technology | - | - |
| Definition: A disorder characteriz | ed by a change in the sound and/o | or speed of the voice. | | | |
| Wheezing | Detectable airway noise with minimal symptoms | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severe respiratory symptoms<br>limiting self care ADL; oxygen<br>therapy or hospitalization<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a high-pitched, whistling sou | ind during breathing. It results from | n the narrowing or obstruction of t | he respiratory airways. | |
| Respiratory, thoracic and mediastinal disorders - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Alopecia | on close inspection; a different hair style may be required to | Hair loss of >=50% normal for<br>that individual that is readily<br>apparent to others; a wig or hair<br>piece is necessary if the patient<br>desires to completely | - | - | - |
| | cover the hair loss but it does<br>not require a wig or hair piece to<br>camouflage | camouflage the hair loss;<br>associated with psychosocial<br>impact | | | |
| Definition: A disorder character | ized by a decrease in density of hair | r compared to normal for a given i | ndividual at a given age and body | location. | |
| Body odor | Mild odor; physician intervention not indicated; self care interventions | Pronounced odor; psychosocial impact; patient seeks medical intervention | - | - | - |
| Definition: A disorder character | ized by an abnormal body smell res | ulting from the growth of bacteria | on the body. | 1 | 1 |
| Bullous dermatitis | Asymptomatic; blisters covering <10% BSA | Blisters covering 10 - 30% BSA;<br>painful blisters; limiting<br>instrumental ADL | Blisters covering >30% BSA;<br>limiting self care ADL | Blisters covering >30% BSA;<br>associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder character | ized by inflammation of the skin cha | racterized by the presence of bull | ae which are filled with fluid. | ı | _ |
| Dry skin | Covering <10% BSA and no associated erythema or pruritus | Covering 10 - 30% BSA and associated with erythema or pruritus; limiting instrumental ADL | Covering >30% BSA and associated with pruritus; limiting self care ADL | - | - |
| Definition: A disorder character | ized by flaky and dull skin; the pores | s are generally fine, the texture is | a papery thin texture. | | _ |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target lesions covering 10 -<br>30% BSA and associated with<br>skin tenderness | Target lesions covering >30%<br>BSA and associated with oral or<br>genital erosions | Target lesions covering >30%<br>BSA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder character | zed by target lesions (a pink-red rin | g around a pale center). | T | 1 | _ |
| Erythroderma | - | Erythema covering >90% BSA without associated symptoms; limiting instrumental ADL | Erythema covering >90% BSA with associated symptoms (e.g., pruritus or tenderness); limiting self care ADL | Erythema covering >90% BSA with associated fluid or electrolyte abnormalities; ICU care or burn unit indicated | Death |
| Definition: A disorder character | zed by generalized inflammatory er | ythema and exfoliation. The inflan | nmatory process involves > 90% o | of the body surface area. | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10 - 30% BSA and associated with erythema or tenderness; limiting instrumental ADL | Covering >30% BSA;<br>associated with erythema or<br>tenderness; limiting self-care<br>ADL | - | - |
| | ized by shrinking of adipose tissue. | <u> </u> | | | |
| Hirsutism | In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | In women, increase in length, thickness or density of hair in a male distribution that requires daily shaving or consistent destructive means of hair removal to camouflage; associated with psychosocial impact | - | - | - |
| Definition: A disorder characteri | ized by the presence of excess hair | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | c and unde |
| androgen control (beard, moust | • • | | | | |
| Hyperhidrosis | Limited to one site (palms, soles, or axillae); self care interventions | Involving >1 site; patient seeks<br>medical intervention; associated<br>with psychosocial impact | Generalized involving sites<br>other than palms, soles, or<br>axillae; associated with<br>electrolyte/hemodynamic<br>imbalance | - | - |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | I | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or<br>density of hair that the patient is<br>either able to camouflage by<br>periodic shaving or removal of<br>hairs or is not concerned | Increase in length, thickness or density of hair at least on the usual exposed areas of the body [face (not limited to beard/moustache area) | - | - | - |
| | enough about the overgrowth to use any form of hair removal | plus/minus arms] that requires<br>frequent shaving or use of<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial | | | |
| Dofinition: A disorder characteri | Zod by hair dansity or langth bayon | impact | a particular body ragion for a part | icular ago or race | ļ |
| Hypohidrosis | zed by hair density or length beyon | Symptomatic; limiting instrumental ADL | Increase in body temperature; | Heat stroke | Death |
| Definition: A disorder characteri | zed by reduced sweating. | | | <b>.</b> | |
| Lipohypertrophy | Asymptomatic and covering <10% BSA | Covering 10 - 30% BSA and associated tenderness; limiting instrumental ADL | Covering >30% BSA and<br>associated tenderness and<br>narcotics or NSAIDs indicated;<br>lipohypertrophy; limiting self<br>care ADL | - | - |
| Definition: A disorder characteri | zed by hypertrophy of the subcutan | eous adipose tissue at the site of | multiple subcutaneous injections of | of insulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by a change in the color of the | nail plate. | T | Τ | 1 |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the<br>nail bed from the nail plate or<br>nail loss; limiting instrumental<br>ADL | - | - | - |
| Definition: A disorder characteri | zed by loss of all or a portion of the | nail. | | | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | - | - | - | - |
| Definition: A disorder characteri | zed by vertical or horizontal ridges | on the nails. | ' | ' | |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder characteri | zed by marked discomfort sensation | n in the skin. | T | Γ | 1 |
| Palmar-plantar<br>erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling, blisters, bleeding, edema, or hyperkeratosis) with pain; limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | - | - |
| | zed by redness, marked discomfort | | | reet. | Т |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance; increased intraocular pressure, glaucoma or retinal hemorrhage; optic neuritis; diuretics indicated; operative intervention indicated | - | - |
| Definition: A disorder characteri | zed by swelling due to an excessive | e accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Painless erythema and<br>erythema covering <10% BSA | Tender erythema covering 10 - 30% BSA | Erythema covering >30% BSA<br>and erythema with blistering;<br>photosensitivity; oral<br>corticosteroid therapy indicated;<br>pain control indicated (e.g.,<br>narcotics or NSAIDs) | Life-threatening consequences; urgent intervention indicated | Death |

| Skin and subcutaneous tissue disorders | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical intervention indicated | Intense or widespread;<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated;<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | - | - |
| Definition: A disorder character | ized by an intense itching sensation | | 1 | I | ' |
| Purpura | Combined area of lesions covering <10% BSA | Combined area of lesions covering 10 - 30% BSA; bleeding with trauma | Combined area of lesions covering >30% BSA; spontaneous bleeding | -<br>Dider lesions are usually a darker | -<br>ourple color |
| and eventually become a browr | | | | , | |
| Rash acneiform | Papules and/or pustules<br>covering <10% BSA, which may<br>or may not be associated with<br>symptoms of pruritus or<br>tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder character | ized by an eruption of papules and p | ,<br>oustules, typically appearing in fac | ce, scalp, upper chest and back. | ' | • |
| Rash maculo-papular | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness) | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruritus,<br>burning, tightness); limiting<br>instrumental ADL | Macules/papules covering<br>>30% BSA with or without<br>associated symptoms; limiting<br>self care ADL | - | - |
| | ized by the presence of macules (fla<br>upper trunk, spreading centripetally | | nown as morbillform rash, it is one | of the most common cutaneous a | dverse |
| Scalp pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | - | - |
| Definition: A disorder character | ized by marked discomfort sensation | n in the skin covering the top and | the back of the head. | Γ | |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA; associated with ulceration | - | - |
| Definition: A disorder character | ized by the degeneration and thinning | ng of the epidermis and dermis. | _ | T | |
| Skin hyperpigmentation | Hyperpigmentation covering <10% BSA; no psychosocial impact | Hyperpigmentation covering >10% BSA; associated psychosocial impact | - | - | - |
| Definition: A disorder character | ized by darkening of the skin due to | excessive melanin deposition. | | | |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | - | - | - |
| Definition: A disorder character | ized by loss of skin pigment. | | | | |
| Skin induration | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to<br>slide or pinch skin; limiting joint<br>movement or orifice (e.g.,<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with signs or symptoms of impaired breathing or feeding | Death |
| | ized by an area of hardness in the s | | T | T | |
| Skin ulceration | Combined area of ulcers <1 cm;<br>nonblanchable erythema of<br>intact skin with associated | Combined area of ulcers 1 - 2 cm; partial thickness skin loss involving skin or subcutaneous | Combined area of ulcers >2 cm;<br>full-thickness skin loss involving<br>damage to or necrosis of | Any size ulcer with extensive destruction, tissue necrosis, or damage to muscle, bone, or | Death |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | - | - | Skin sloughing covering <10%<br>BSA with associated signs (e.g.,<br>erythema, purpura, epidermal<br>detachment and mucous<br>membrane detachment) | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>epidermal detachment and<br>mucous membrane<br>detachment) | Death |
| Definition: A disorder characterize | ed by less than 10% total body ski | n area separation of dermis. The | syndrome is thought to be a hyper | sensitivity complex affecting the s | kin and the |
| mucous membranes. | Г | Γ | Γ | Γ | 1 |
| Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | - | - | - |
| Definition: A disorder characterize | ed by local dilatation of small vess | els resulting in red discoloration o | f the skin or mucous membranes. | | |
| Toxic epidermal necrolysis | - | - | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| Definition: A disorder characterize mucous membranes. | ed by greater than 30% total body | skin area separation of dermis. T | he syndrome is thought to be a hy | persensitivity complex affecting th | e skin and the |
| Urticaria | Urticarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 - 30% BSA; oral intervention indicated | Urticarial lesions covering >30%<br>BSA; IV intervention indicated | - | - |
| Definition: A disorder characterize | ed by an itchy skin eruption charac | cterized by wheals with pale interi | ors and well-defined red margins. | | |
| Skin and subcutaneous tissue disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| Social circumstances | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Menopause | Menopause occurring at age 46 - 53 years of age | Menopause occurring at age 40 - 45 years of age | Menopause occurring before age 40 years of age | - | - |
| Definition: A disorder characteriz | ed by the permanent cessation of | menses, usually defined by 12 co | nsecutive months of amenorrhea i | n a woman over 45 years of age. | |
| Social circumstances - Other, specify | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |
| | | | disabling; limiting self care ADL | | |

| Surgical and medical procedures | | | | | |
|---|---|---|---|---|---|
| | | Grade | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Surgical and medical | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| procedures - Other, specify | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent intervention indicated | |
| | observations only; intervention | indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| 1 | | | disabling; limiting self care ADL | | |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Capillary leak syndrome | - | Symptomatic; medical intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by leakage of intravascular flui<br>ck syndromes, low-flow states, ische | · | • | • | |
| Flushing | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Symptomatic, associated with hypotension and/or tachycardia; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by episodic reddening of the fa | ice. | İ | 1 | |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a localized collection of bloo | od, usually clotted, in an organ, sp | ace, or tissue, due to a break in th | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by an uncomfortable and temp | orary sensation of intense body w | armth, flushing, sometimes accom | panied by sweating upon cooling. | |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic<br>BP 140 - 159 mm Hg or<br>diastolic BP 90 - 99 mm Hg);<br>medical intervention indicated;<br>recurrent or persistent (>=24<br>hrrs); symptomatic increase by<br>>20 mm Hg (diastolic) or to<br>>140/90 mm Hg if previously | Stage 2 hypertension (systolic<br>BP >=160 mm Hg or diastolic<br>BP >=100 mm Hg); medical<br>intervention indicated; more<br>than one drug or more intensive<br>therapy than previously used<br>indicated<br>Pediatric: Same as adult | Life-threatening consequences<br>(e.g., malignant hypertension,<br>transient or permanent<br>neurologic deficit, hypertensive<br>crisis); urgent intervention<br>indicated<br>Pediatric: Same as adult | Death |
| Definition: A disorder characte | rized by a pathological increase in b | WNL; monotherapy indicated<br>Pediatric: recurrent or persistent<br>(>=24 hrs) BP >ULN;<br>monotherapy indicated | | ng 140 over 90 mm Hg. | |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention or hospitalization indicated | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder characte | rized by a blood pressure that is belo | ow the normal expected for an ind | ividual in a given environment. | | |
| Lymph leakage | - | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by the loss of lymph fluid into t | he surrounding tissue or body cav | ity. | 1 | |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery skin texture; papillary formation; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A disorder characte | erized by excessive fluid collection in | tissues that causes swelling. | | | |
| Lymphocele | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | - | - |
| Definition: A disorder characte | erized by a cystic lesion containing ly | mph. | 1 | | |
| Peripheral ischemia | - | Brief (<24 hrs) episode of ischemia managed non-<br>surgically and without permanent deficit | Recurring or prolonged (>=24<br>hrs) and/or invasive intervention<br>indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by impaired circulation to an ex | ktremity. | 1 | | |
| Phlebitis | - | Present | - | - | - |
| Definition: A disorder characte | rized by inflammation of the wall of a | vein. | | | |
| Superficial thrombophlebitis | - | Present | - | - | - |
| Definition: A disorder characte | erized by a blood clot and inflammation | on involving a superficial vein of th | e extremities. | | |

| | | Vascular disord | ers | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Superior vena cava syndrome | Asymptomatic; incidental finding of SVC thrombosis | Symptomatic; medical intervention indicated (e.g., anticoagulation, radiation or chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting) | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery) | Death |
| | ed by obstruction of the blood flow | in the superior vena cava. Signs | and symptoms include swelling ar | nd cyanosis of the face, neck, and | upper arms, |
| cough, orthopnea and headache Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | Thrombosis (e.g., uncomplicated pulmonary embolism [venous], non-embolic cardiac mural [arterial] thrombus), medical intervention indicated | Life-threatening (e.g., pulmonary embolism, cerebrovascular event, arterial insufficiency); hemodynamic or neurologic instability; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream. | Т | 1 |
| Vasculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of peripheral or visceral ischemia; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the w | rall of a vessel. | | | |
| Visceral arterial ischemia | - | Brief (<24 hrs) episode of ischemia managed medically and without permanent deficit | Prolonged (>=24 hrs) or recurring symptoms and/or invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a decrease in blood supply | due to narrowing or blockage of a | visceral (mesenteric) artery. | | |
| Vascular disorders - Other,<br>specify | 1 , 1 , | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |







NIH Publication No. 09-5410 Revised June 2010 Reprinted June 2010



### APPENDIX 2. PEMPHIGUS DISEASE AREA INDEX (PDAI)

#### Pemphigus Disease Area Index (PDAI)

| Skin | Activity | | Damage |
|---|---|---|---|
| Anatomical Locatio | Erosion/Blisters or new erythem | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion | |
| | 0 absent 1 1-3 lesions, up to one >2 cm in any diameter, none > 6 cm 2 2-3 lesions, at least two > 2 cm diameter, none > 6 cm 3 >3 lesions, none > 6 cm diameter 5 >3 lesions, and/or at least one >6 cm 10 >3 lesions, and/or at least one lesion >16 cm diameter or entire area | Number<br>lesions if<br>≤ 3 | 0 absent<br>1 present |
| Ears | | | |
| Nose | | | |
| Rest of the face | | | |
| Neck | | | |
| Chest | | | |
| Abdomen | | | |
| Back, buttocks | | | |
| Arms | | | |
| Hands | | | <u> </u> |
| Legs | | | |
| Feet | | | |
| Genitals | | | |
| Total skin | /120 | | /12 |
| Scalp | | | |
| Scalp | Erosion/Blisters or new erythem | Post-inflammatory<br>hyperpigmentation or erythema<br>from resolving lesion | |
| | 0 absent 1 in one quadrant 2 two quadrants 3 three quadrants 4 affects whole skull 10 at least one lesion > 6 cm | 0 absent<br>1 present | |
| Total Scalp (0-10) | /10 | | /1 |
| Mucous men | nbrane | | |
| Anatomical | Erosion/Blisters | | |
| Location | 0 absent<br>1 1 lesion<br>2 2-3 lesions<br>5 > 3 lesions or 2 lesions > 2 cm<br>10 entire area | Number<br>lesions<br>if ≤ 3 | |
| Eyes | | | |
| Nose | | | |
| Buccal mucosa | | | |
| Hard palate | | | |
| Soft palate | | | |
| Upper gingiva | | | |
| Lower gingiva | | | |
| Tongue | | | |
| Floor of mouth | | | |
| Labial bucosa | | | |
| Posterior pharynx | | | |
| | | | I |
| Anogenital | | - | l . |

Copyright ©2007 University of Pennsylvania; All Rights Reserved.

# APPENDIX 3. AUTOIMMUNE BULLOUS DISEASE QUALITY OF LIFE (ABQOL) QUESTIONNAIRE

 Syntimmune, Inc.

### **ABQOL Questionnaire**

| Name: | Date: |
|---|---|
| DOB: Sex: M/F | Contact Number: |
| Pemphigus Subtype: Pemphigus Vulgaris | <ul> <li>Epidermolysis Bullosa Aquisita</li> </ul> |
| □ Bullous Pemphigoid | □ Linear IgA Bullous Dermatoses |
| □ Pemphigus Follaceus | □ Mucous Membrane Pemphigoid |
| □ Other | · |
| The following questions ask about the ways in quality of life. | which <i>blistering disease treatments</i> affect your |
| Please choose an option from the right hand co felt within the last week. | olumn which most closely correlates to how you |
| Please time your survey in minutes and se | conds – start time AM/PM |
| <ol> <li>In regards to your blistering disease,<br/>does your skin burn, sting or hurt in</li> </ol> | All the time Sometimes |
| any way? | Occasionally Not at all |
| 2. In regards to your blistering disease, | All the time |
| does your skin itch? | <ul><li>Sometimes</li><li>Occasionally</li></ul> |
| | Not at all |
| Have you had to change your clothing because of your blictoring | I have to be very careful with how tight my elething is and what materials they |
| clothing because of your blistering disease? | my clothing is and what materials they<br>are made of – I have had to change what<br>I wear all the time |
| | I have had to change most of the things I wear |
| | I have had to change some of the things I wear |
| | I have never had to change what I wear |
| 4. Do you notice your skin heals slowly? | I notice this all the time I notice this sometimes |
| | I notice this occasionally |
| Do you have difficulty bathing or | |
| showering because of your blistering | o Sometimes |
| disease? | Occasionally Not at all |

| In regards to your blistering disease,<br>does your mouth have erosions<br>which are painful? | <ul><li> All the time</li><li> Sometimes</li><li> Occasionally</li><li> Not at all</li></ul> |
|---|---|
| In regards to your blistering disease, do your gums bleed easily? | <ul><li> All the time</li><li> Sometimes</li><li> Occasionally</li><li> Not at all</li></ul> |
| Does your blistering disease results in you having to avoid food or drinks that you enjoy? | I can no longer eat any of the foods I used to enjoy I can eat some of the foods I enjoy I can eat most of the foods I enjoy I can eat anything I like |
| 9. As a result of your blistering disease, are you embarrassed about your appearance? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 10. Do you feel depressed or angry because of your blistering disease? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 11. Do you feel anxious or cannot relax as a result of your blistering disease? | <ul><li>All the time</li><li>Sometimes</li><li>Occasionally</li><li>Not at all</li></ul> |
| 12. Do you worry that friends and family find your blistering skin condition tiresome? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 13. Is your blistering disease causing sexual difficulties? | <ul> <li>All the time</li> <li>Sometimes</li> <li>Occasionally</li> <li>Not at all</li> </ul> |
| 14. Does your blistering disease affect relationships with friends or loved ones? | <ul> <li>I have had to end a relationship because of my disease OR I cannot have a relationship because of my disease</li> <li>Relationships are very difficult</li> <li>Relationships are a little difficult</li> <li>This has not affected my relationships</li> </ul> |

| 15. Does your blistering disease affect your social life? | <ul> <li>I cannot go out to socialize any more</li> <li>I can only go to some social events</li> <li>I can go to most social events</li> <li>My social life is not affected</li> </ul> |
|---|---|
| 16. Does your blistering disease affect your work or study? | <ul> <li>Yes, I can no longer work or study</li> <li>Yes, I find it difficult to work or study</li> <li>Yes, it is a little harder than before to work or study</li> <li>No, I am not affected OR not applicable (N/A)</li> </ul> |
| 17. Do employers discriminate against you because of your blistering disease? | I cannot find a job due to my blistering disease I have had to change jobs due to my blistering disease I still have my job but it is more difficult than before My employers are completely understanding OR not applicable (N/A) |

Please indicate the time taken to finish the survery: minutes seconds

Thank you for taking the time to complete this questionnaire

#### APPENDIX 4. SKINDEX-29

 Syntimmune, Inc.

# **DERMATOLOGY SURVEY**

This survey concerns the skin condition which has bothered you the most during the past four weeks.

These questions concern your feelings over the past 4 weeks about **the skin condition that has bothered you the most**. Check the answer that comes closest to the way you have been feeling.

| HOW OFTEN DURING THE PAST FOUR WEEKS DO THESE STATEMENTS DESCRIBE YOU? | NEVER | RARELY | SOMETIMES | OFTEN | ALL THE<br>TIME |
|---|---|---|---|---|---|
| 1. My skin hurts | 1 | $\square_2$ | Пз | □4 | □5 |
| 2. My skin condition affects how well I sleep | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 3. I worry that my skin condition may be serious | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 4. My skin condition makes it hard to work or do hobbies | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 5. My skin condition affects my social life | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 6. My skin condition makes me feel depressed | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 7. My skin condition burns or stings | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 8. I tend to stay at home because of my skin condition | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 9. I worry about getting scars from my skin condition | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 10. My skin itches | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 11. My skin condition affects how close I can be with those I love . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 12. I am ashamed of my skin condition | $\square_1$ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 13. I worry that my skin condition may get worse | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 14. I tend to do things by myself because of my skin condition . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 15. I am angry about my skin condition | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 16. Water bothers my skin condition (bathing, washing hands) . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 17. My skin condition makes showing affection difficult | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 18. I worry about side-effects from skin medications / treatments . | $\square_1$ | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 19. My skin is irritated | □1 | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 20. My skin condition affects my interactions with others | □1 | $\square_2$ | $\square_3$ | $\square_4$ | □5 |

Please turn to next page

These questions concern your feelings over the past 4 week about **the skin condition that has bothered you the most**. Check the answer that comes closest to the way you have been feeling.

| HOW OFTEN DURING THE PAST 4 WEEK DO THESE STATEMENTS DESCRIBE YOU? | NEVER | RARELY | SOMETIMES | OFTEN | ALL THE<br>TIME |
|---|---|---|---|---|---|
| 21. I am embarrassed by my skin condition | <b>□</b> 1 | $\square_2$ | □3 | □4 | $\square_5$ |
| 22. My skin condition is a problem for the people I love | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 23. I am frustrated by my skin condition | □1 | $\square_2$ | □₃ | $\square_4$ | $\square_5$ |
| 24. My skin is sensitive | □1 | $\square_2$ | Пз | $\square_4$ | $\square_5$ |
| 25. My skin condition affects my desire to be with people | □1 | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 26. I am humiliated by my skin condition | □1 | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 27. My skin condition bleeds | □₁ | $\square_2$ | $\square_3$ | $\square_4$ | $\square_5$ |
| 28. I am annoyed by my skin condition | □1 | $\square_2$ | $\square_3$ | □4 | $\square_5$ |
| 29. My skin condition interferes with my sex life | □1 | $\square_2$ | $\square_3$ | $\square_4$ | □5 |
| 30. My skin condition makes me tired | □₁ | $\square_2$ | □₃ | $\square_4$ | □5 |

#### APPENDIX 5. COHORT 2 ALTERNATE SCHEDULE OF EVENTS TABLE

 Syntimmune, Inc.

Table 10. Study Assessments for Cohort 2 (Alternate Weekly Dosing Option)

| | Screening | Loa | ading | | | | | | Mair | itenanc | e | | | | F | ollow-U | Ú <b>p</b> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 |
| Time Point<br>(Study Day) | -14 to -1 | 0<br>Baseline | 7<br>(±1 d) | 14<br>(±1 d) | 21<br>(±3 d) | 28<br>(±3 d) | 35<br>(±3 d) | 42<br>(±3 d) | 49<br>(±3 d) | 56<br>(±3 d) | 63<br>(±3 d) | 70<br>(±3 d) | 77<br>(±3 d) | 84<br>(±3 d) | 91<br>(±5 d)<br>or ET<br>Visit | 112<br>(±5 d) | 140<br>(±5 d)<br>EOS<br>Visit |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Demographics/medical history | X | | | | | | | | | | | | | | | | |
| Inclusion/exclusion | X | | | | | | | | | | | | | | | | |
| Physical examination <sup>a</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pulse oximetry <sup>c</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Clinical safety labs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy test <sup>e</sup> | X | X | | | X | | | | | | | | | | X | | X |
| Hepatitis and HIV screen | X | | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>f</sup> | X | X | | X | X | | | | | | | | | | X | | X |
| Tetanus and VZV antibodies <sup>g</sup> | | X | | | X | | | | | | | | | | X | | X |
| PDAI <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PK sampling <sup>i</sup> | | X | X | X | X | | X | | | | | | | X | | | |
| Immunogenicity <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Study drug administration <sup>k</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG1-4) <sup>l</sup> | X | X | X | Х | Х | Х | X | X | X | Х | X | X | X | X | X | X | $X^q$ |
| CIC | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Anti-Dsg (1 and 3) antibody titers | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| C3 and AECA <sup>m</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| FCGR2A by buccal swab <sup>n</sup> | | X | | | | | | | | | | | | | | | |
| RNA sequencing | | X | | | X | | | | | | | | | | X | | |
| Immunophenotyping° | | X | | | X | | | | | | | | | | X | | |
| Exploratory pemphigus immune response biomarkers | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

 Syntimmune, Inc.

| Photography <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HR-QoL assessments | X | | | X | | | | | | | | | | X | | X |
| Adverse events | To be collected from the date that the ICF is signed through the last study visit | | | | | | | | | | | | | | | |
| Concomitant medications | To be collected from within 14 days prior to Day 0 through the last study visit | | | | | | | | | | | | | | | |

CIC = circulating immune complexes; d = day(s); ECG = electrocardiogram; EOS = end of study; ET= early termination; FCGR2A = Fc gamma R2a receptor; HIV = human immunodeficiency virus; HR-QoL = health-related quality of life; ICF = informed consent form; Ig = immunoglobulin; PDAI = Pemphigus Disease Area Index; PK = pharmacokinetic; VZV = varicella-zoster virus

- a. Complete physical examination, including weight, to be performed. Height and body mass index will be additional assessments conducted at screening only.
- b. **Vital sign** measurements (sitting blood pressure, heart rate, respiratory rate, and oral temperature) to be obtained after 5 minutes of seated rest. Any abnormal measurements are to be repeated after 5 minutes of rest. Vital sign measurements will be taken on all study visits. On dosing days, vital sign measurements will be collected immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour and 2 hours following completion of the infusion.
- c. **Pulse oximetry:** On dosing days, pulse oximetry to be measured immediately prior to the infusion; 15, 30, and 45 minutes after the start of the infusion; at completion of the infusion; and 30 minutes, 1 hour, and 2 hours following completion of the infusion.
- d. Clinical safety labs: hematology, clinical chemistry, and urinalysis. See Section 7.5 for a complete list. Full clinical safety lab draws will be collected at screening and at all study visits prior to infusion if applicable.
- e. **Pregnancy test (women of childbearing potential only):** To be performed at time of screening and prior to dose on dosing days if applicable. Urine or serum test is acceptable; however, positive urine tests must be confirmed with serum testing.
- f. Digital 12-lead ECG to be obtained after 5 minutes of rest in the supine position and in triplicate approximately 1 minute apart. See Section 7.6 for additional information. On dosing days, to be obtained approximately 5 minutes after the completion of infusion.
- g. **Serology:** Any subject whose baseline value for tetanus or VZV was above the protective level at baseline and is not within 30% of the baseline value or is below the protective level by End of Follow-up, will be referred to their primary care physician for further management. See Section 7.5.3 for additional information.
- h. PDAI will be administered at screening. Subject eligibility requires a PDAI total activity score >4. Thereafter, assuming eligibility, the PDAI will be administered during Treatment Period and Follow-up Period. See Section 7.7 for additional information.
- i. **PK:** On dosing days if applicable, serum samples will be collected just prior to the start of study drug infusion (pre-dose) and at 5 minutes, 1 and 2 hours after the end of study drug infusion. See Section 7.5.4 for additional information.
- j. Immunogenicity: Samples will be collected pre-dose when collected on dosing days. See Section 7.5.6 for additional information.
- k. Prior to **study drug infusion**, SYNT001 drug product is to be diluted in dextrose 5% in water to a total volume of 250 mL and administered intravenously over 1 hour ±15 minutes using a 0.2-micron, inline filter. See Section 4 for additional information.
- 1. Immunoglobulins (IgG, IgA, IgM) and IgG subtypes (IgG 1-4): Collected for measurements of IgG, IgG subtypes (IgG1-4), IgA, and IgM at every visit. On dosing days, samples are collected prior to infusion of study drug. See Section 7.5.5 for additional information.
- m. Exploratory pharmacodynamic samples (C3 and AECA): Collected pre-dose when collected on dosing days. See Section 7.5.5 for complete information.
- n. Buccal samples to be collected pre-dose.
- o. **Immunophenotyping** by flow cytometry for measurement of CD3<sup>+</sup>CD4<sup>+</sup> T, CD3<sup>+</sup>CD8<sup>+</sup> T, monocytes, natural killer (NK) cells, and B cells. Collect samples pre-dose on dosing days.
- p Photographs of all active lesions taken pre-dose on dosing days. Subjects who begin a steroid taper will have additional photographs taken at the clinic visit during which the decision to begin the taper is made.
- q Subjects whose total IgG is not within 30% of their Day 0 baseline value and not above 500 mg/dL at Day 140 will be referred for further management.

 Syntimmune, Inc.

## PROTOCOL AMENDMENT **SUMMARY OF CHANGES**

**Protocol Title:** A Phase 1b/2, Multicenter, Open-Label, Safety, and Dose-Finding Study of

SYNT001 in Subjects with Pemphigus (Vulgaris or Foliaceus)

**Protocol Number:** SYNT001-103

**Study Drug:** SYNT001

**Sponsor:** Syntimmune, Inc.

116 Huntington Avenue

Suite 301

Boston, MA 02116

PPD **Medical Monitor:** 

Wallace House

17-21 Maxwell Place Stirling, Scotland FK81JU

Mobile Phone: PPD

ext. PPD Office Phone: PPD

**Original Protocol:** 18 January 2017 21 March 2017 **Amendment 1.0:** Amendment 2.0 12 April 2017 Amendment 3.0 10 October 2017 Amendment 4.0 08 June 2018

Amendment 5.0 18 September 2018

#### **CONFIDENTIALITY STATEMENT**

This document is the property of Syntimmune, Inc. This document contains confidential information, which should not be copied, referred to, released, or published without written approval from Syntimmune. Investigators are cautioned that the information given in this brochure might be subject to change and revision. Any conclusion regarding efficacy and safety must be considered provisional.

#### BACKGROUND

Protocol amendment Version 5.0 of the SYNT001-103 protocol was issued on 18 September 2018.

Syntimmune is amending the SYNT001-103 protocol to adjust the dosing schedule and cohort options. Because enrollment in Cohort 1 is complete, subjects will be enrolled in Cohort 2 which will now evaluate 3 weekly loading doses followed by 5 every other week maintenance doses, with the option to adjust to weekly dosing, if needed. Most updates in the amendment were incorporated to reflect this change, as well as refine how the ongoing safety of subjects in Cohort 2 would be monitored. The number of sites was increased to aid in enrollment and PDAI and photography assessments are now included at every post-treatment visit for Cohort 2 to better assess efficacy. PDAI also assessment added at screening for Cohort 2.

General grammatical, typographical, and formatting updates have been made throughout the document to provide consistency and clarity, reduce redundancy, and improve readability. These changes are not detailed in the summary below. Please see Amendment 5 for details.

#### **SUMMARY OF CHANGES**

With this update, the following changes since Version 4.0 have been made:

Table 1. Summary of Changes: Protocol Version 5.0

| Section Number and Title | Description of Change |
|---|---|
| Sponsor<br>Signature | The name of the Sponsor Representative has been updated. |
| Section 1,<br>Protocol Synopsis | Below is a summary of changes to the protocol synopsis; refer to the changes described for the individual protocol sections for more detail: • Increased the number of study sites from 10 to 20 global sites to support subject enrollment. |
| | Study objectives and endpoints were updated to reflect changes to the dosing regimen (every other week in maintenance phase), to clarify that serum is used for pharmacokinetic analyses, and to update how analysis summaries will be presented. |
| | <ul> <li>The Study design and Methodology sections have been merged.</li> <li>The Study design not only describes changes to cohorts but also includes the role of the Dose Escalation Committee (DEC), Sponsor Medical Lead, and stopping and dose escalation rules.</li> </ul> |
| | • The Number of subjects section has been updated to reflect the changes in the number of subjects and that Cohort 1 may enroll "up to" 8 subjects and Cohort 2 may enroll "up to" 12 subjects. |
| | The Study population section was modified to better define the population. |
| | • Inclusion criterion #4a was updated to reduce the last previous dose of rituximab or other anti-CD20 monoclonal antibodies from >12 months to >9 months prior to screening. |
| | • Inclusion criterion #9 was updated to reflect that male subjects are only required to use contraception through the final study visit. |
| | <ul> <li>Exclusion criterion #12 was updated to specify "at screening."</li> <li>Additional detail regarding dose/cohort changes has been added to Study drug, dosage, and administration and Duration of subject participation sections.</li> </ul> |
| | More detail was added for clarity regarding corticosteroids. |
| | • In the statistical consideration section, analyses have been updated to reflect changes to the dosing regimen (every other week in maintenance phase) and to update how analysis summaries will be presented. |
| Study Diagram | Study Diagram has been added for clarity around the changes to study design and the reduction in the number of cohorts to 2. |

| | • Cohort 2 has been modified to 3 weekly loading doses of 30 mg/kg followed by 5 every other week doses of 10 mg/kg and the number of subjects enrolled will be up to 12. |
|---|---|
| | The original Cohort 2 and optional Cohort 4 were removed. |
| | • The Sponsor Medical Team will conduct the 24-hour and 7-day safety reviews for subjects in Cohort 2. |
| | • Ongoing safety review may result in may modified dosing regimen (e.g. 10 weekly maintenance doses at 10-30 mg/kg). |
| Schedule of<br>Events | Tables 3 and 4 (original Cohort 2 and Cohort 3) were deleted. |
| | Table 3 (Cohort 2): This table reflects a new dosing schedule with loading and maintenance doses, as well as the increase of PDAI and photography assessments to every post-treatment visit. PDAI also added at screening. See Table 3 for details. |
| List of Abbreviations | The table was updated to include all abbreviations throughout the synopsis and protocol text. Each abbreviation was defined the first time used in both the synopsis and protocol text. |
| Section 2, | Background and Rationale |
| Background and Rationale | Text has been added to describe SYNT001's predicted mechanism of action |
| | Additional indications identified as IgG-mediated autoimmune disorders have been removed |
| | Selection of Doses in this Study |
| | Details of mathematical modeling of study dose selection were added. |
| | Details of non-clinical and clinical studies supporting the proposed<br>Cohort 2 dose and dosing regimen were added. |
| Section 3, Study<br>Objectives and<br>Endpoints | • Study objectives and endpoints were updated to reflect changes to the dosing regimen (every other week in maintenance phase), to clarify that serum is used for pharmacokinetic analyses, and to update how analysis summaries will be presented. |
| Section 4, Study | <ul> <li>The secondary objectives were reordered to reflect their importance.</li> <li>Description of SYNT001</li> </ul> |
| Drug | Added that Investigators are allowed to adjust the duration of the infusion to increase tolerability up to 4 hours, if needed. |
| | <ul> <li>Dose Requirements</li> <li>It has been clarified that subject doses will be limited to 5000 mg. A subject with a body weight that extrapolates to a dose &gt; 5000 mg, will only receive 5000 mg.</li> </ul> |
| Section 5, Study | The number of study sites was increased from 10 to 20. |
| Design | The study design has been updated to reflect changes in dosing regimen for Cohort 2. |
| | • Cohort 1 number of subjects has been modified from 8 to <u>up to</u> 8. |

| | • Cohort 2 has been modified to 3 weekly loading doses of 30 mg/kg followed by 5 every other week doses of 10 mg/kg and the number of subjects enrolled will be up to 12. |
|---|---|
| | Original Cohort 2 and optional Cohort 3 were removed. |
| | • The Sponsor Medical Team will conduct the 24-hour and 7-day safety reviews for Cohort 2. |
| | • Ongoing safety review may result in may modified dosing regimen (e.g. 10 weekly maintenance doses at 10-30 mg/kg). |
| | • Duration of Subject Participation was added to the body of the protocol for consistency with the synopsis. |
| Section 6, Study<br>Population | <ul> <li>Target Population</li> <li>Based on the new study design, the total number of subjects has been changed to a maximum of 20 subjects, but the number is not included in this section, just a description of the study population.</li> <li>Inclusion Criteria</li> </ul> |
| | • Inclusion criterion #4a was updated to reduce the last previous dose of rituximab or other anti-CD20 monoclonal antibodies from >12 months to >9 months prior to screening. |
| | • Inclusion criterion #9 was updated to reflect that male subjects are only required to use contraception through the final study visit. |
| | Exclusion Criteria |
| ~ ~ . | • Exclusion criterion #12 was updated to specify "at screening." |
| Section 7, Study<br>Procedures | • References to specific days have been removed because of the addition of the separate Cohort 2 table and possibility of following the optional weekly schedule in Appendix 3. |
| | • Virology assessments were removed from Table 6 because they are not included with clinical laboratory panels. |
| | • PK parameters studied in Cohort 1 differ from (the) successive cohort(s) and which include maximum serum concentration of SYNT001 and the associated T <sub>max</sub> . |
| | • Pharmacodynamic Assessment (Table 7) has been updated to include timing of testing for Cohort 2 |
| | A subsection re: corticosteroid use was added for clarity. |
| Section 8, Study<br>Assessments | Sections were edited to reflect the updates to assessments performed in the new schedule of events for Cohort 2. See Section 8 for details. |
| Section 9, Study | Subject Withdrawal |
| Rules | Details were added to distinguish between follow up assessments for |
| | subjects who prematurely discontinue study drug versus subjects who |
| | <ul> <li>prematurely discontinue from the study.</li> <li>Details were added to specify which study visits the subject should be encouraged to attend in each case above.</li> </ul> |
| | Stopping Rules |

| Τ | |
|---|---|
| | • The description of dose escalation stopping rules now reflects that Cohort 2 will not be a dose escalation cohort. |
| | <ul> <li>Decisions regarding study stopping rules originally to be made by the<br/>DEC were updated to be decided by the Sponsor Medical Lead.</li> </ul> |
| Section 10, | No substantial changes were made to this section; only updates to |
| Evaluation of | abbreviations and minor corrections for consistency. |
| Safety | Warnings and Precautions |
| | • Allowed vaccinations were updated to 28 days after the final dose of |
| | study drug rather than discretion of investigator. |
| Section 11, | "Data" was updated to "analysis" in headings. |
| Statistical | Details of analyses have been updated to reflect changes to the dosing |
| Considerations | regimen (every other week in maintenance phase) and to update how |
| | analysis summaries will be presented. |
| | Safety Analysis |
| | <ul> <li>More detail was added to the safety analyses to be performed.</li> </ul> |
| | • Relationship of adverse events (AEs) to study drug was defined as in |
| | the AE section (related/not related). |
| | • The lab analyses were updated to be formed by a central laboratory. |
| | Pharmacokinetic Analysis |
| | PK and PD analyses were moved to separate sections. |
| | • Details were made more general to cover different analyses performed in the 2 cohorts. |
| | Pharmacodynamic (PD) Analysis |
| | Details of the presentation of disease activity marker results were |
| | added. |
| Sections 12-14 | No edits other than global changes mentioned below. |
| Appendix 5 | Appendix was added to include an alternate schedule of events for |
| G1.1.1.61 | Cohort 2 (weekly dosing) |
| Global Changes | • Edits and formatting changes have been made throughout to improve clarity and readability. |
| | • Typographical and formatting corrections as well as corrections for consistency have been made. |